







#### **Clinical Study Protocol**

Drug Substance Olaparib (AZD2281)

Study Code D081CC00006

Study Number BIG 6-13, NSABP B-55

5 Version

Date 18 May 2018

A randomised, double-blind, parallel group, placebo-controlled multi-centre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline BRCA1/2 mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy

Sponsor: AstraZeneca AB, 151 85 Södertälje, Sweden

Clinical Study Protocol Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5

Date 18 May 2018

#### VERSION HISTORY

#### Version 5, 18 May 2018

The primary reason for this protocol amendment is to revise the sample size of the study. In addition, revisions have been made to align with current practice, safety updates and to clarify procedures. Minor editorial changes have also been made but are not included in this summary table.

Statistical background - Rationale for amendment:

To support the addition of the ER+ cohort in protocol version 4 a simulation study was undertaken with the objective to predict accrual of events and therefore the timing of the interim and primary analyses. The simulation study included relevant operating characteristics for the anticipated possible proportions enrolled in each of the 4 subgroups, survival was modelled by piecewise exponential distribution for which annualised hazard according to the respective subgroups were taken from the most recent published data (Dent et al 2007, Cortazar et al 2014, Swain et al 2013).

Following the observation of lower than anticipated event rate (using data extracted on 25 August 2017), it was clear that the published data used for the simulations were too pessimistic with respect to event rates for the Triple negative adjuvant population that have been recruited into Study D081CC00006 (OlympiA) since 2014.

Further predictions were run using the current data (extract date 10 November 2017) and applying AstraZeneca's 'Shiny' oncology event prediction R package. A survival model assuming a Weibull distribution was fitted to the previous study data and used to predict future survival times. Whilst the simulation study simulated over varying proportions enrolled in each sub group, by using the current data, the predictions were based on 1153 patients of whom 15% were ER+ and the ratio of Adjuvant to Neoadjuvant was roughly 1:1. An 8% drop-out rate for the first 12 months, not previously included, was incorporated based on the rate observed so far. The programme forecasted future enrolment from 1153 to 1800 based on the recent observed enrolment rate. There was also no need to adjust this forecast for delays in enrolment due to the protocol amendment.

Given the predictions for timing of the interim and primary analysis it was decided to increase the sample size to 1800 and for the power to remain at 90%. Because the event rate was lower than anticipated, the restriction to have a minimum 2 year follow-up after the last patient enrolled could be removed. Patient enrolment would continue about one year longer than originally anticipated and more patients would be enrolled, thus providing an increase in the number of patient years of follow-up at the time of primary analysis even without the 2 year minimum follow-up criterion.

| Applicable section number(s)/title | Nature of revision |
|---|---|
| Title page | Inclusion of Merck logo. |
| List of olympia protocol authors | List of authors updated. |
| Protocol synopsis 3.2.3 Study Population 12.2.2 Analysis of secondary endpoints 12.2.7 Sample size justification | Number of patients planned has been increased from 1500 to 1800. Number of centres increased from 500 to 700. |
| Protocol synopsis 12.2.7 Sample size justification | The estimation for study recruitment has been increased to 5 years (previously 4.5 years) to account for the 300 extra patients. |
| Protocol synopsis 6.2.5 Patient management post-primary analysis 12.2.1.1 Primary analysis 12.2.2 Analysis of secondary endpoints 12.2.7 Sample size justification | Removed minimum 24 month follow-up from the data cut-off from the primary analysis as the expected high event rate in the first 2 years has not been seen. |
| Protocol synopsis 12.1.1 Full analysis set 12.2.6 Interim analysis | Interim analysis will now be triggered by events in the first 900 patients (previously 750 patients). |
| 1.1.9.1 Olaparib monotherapy studies in breast cancer patients | Addition of efficacy data for Study D0819C00003 (OlympiAD). |
| 1.4 Benefit/risk and ethical assessment | Addition of details (to the potential benefit section) for the olaparib tablet formulation approval for patients with deleterious or suspected deleterious <i>gBRCAm</i> , HER2-negative metastatic breast cancer. |
| 3.1 Overall study design, flow chart and study schedules 3.2.1 Rationale for study design 6.2.2 On-treatment assessments | Text regarding mammogram and/or breast MRI scans amended to include ipsilateral and/or contralateral scanning. Clarification provided regarding the use of ultrasound in patients who underwent a bilateral mastectomy and for male patients. |
| <ul><li>6.2.3 Efficacy follow-up assessments</li><li>6.3.1 Tumour evaluation</li></ul> | |

| Applicable section number(s)/title | Nature of revision |
|---|---|
| 3.1 Overall study design, flow chart and study schedules | Information added to Table 3 footnote to clarify monitoring of all ongoing AEs/SAEs and any new AEs/SAEs identified during the 30 calendar days. |
| | Pneumonitis included in the events occurring after the 30 day follow-up period that should be reported as an SAE. |
| 3.1 Overall study design, flow chart and study schedules 6.2.1 Screening procedures 6.2.2 On-treatment assessments 6.4.9.1 Serum or urine pregnancy test | Timings for pregnancy testing in women of childbearing potential clarified. Pregnancy tests on blood or urine amended to serum or urine. |
| 4.1 Inclusion criteria | Criterion 11B: Methods of contraception text amended. |
| 4.2 Exclusion criteria | Criterion 11: Use of strong and moderate CYP3A inhibitors text amended and new criteria included to cover the use of concomitant strong and moderate CYP3A inducers on study. |
| | Criterion 13: Criteria modified to patients with current or past history of haematologic malignancies and any clonal non-malignant haematological disorder which predisposes the patient to develop a haematological malignancy. |
| 5.1.1 Meals and dietary restrictions | New section to cover that grapefruit juice consumption on study is prohibited. |
| 5.1.2 Contraception Appendix E | Text updated to specify two highly effective forms of contraception should be used in combination and this should be started from the signing of the informed consent. Male patient contraception text clarified. |
| 5.4.2 Methods for unblinding individual patients | Text revised to include post treatment data verification for unblinded patients. |

| Applicable section number(s)/title | Nature of revision |
|---|---|
| 5.5 Treatments | Table 5 and Table 6 updated to include temporary dose reductions to 300 and 200 mg due to CYP3A inhibitor exposure. Table 8 and Table 9 added to cover dose reductions for management of renal impairment and the use of strong or moderate CYP3A inhibitors while on study. |
| 5.5.6.3 Renal impairment | New section to cover management of renal impairment while on study. |
| 5.5.6.7 Interruptions for intercurrent non-toxicity related events | Additional text provided advising caution while driving or using machinery in case of AEs of asthenia, fatigue and dizziness. |
| 5.6.2 Restricted concomitant medications | Section name changed from CYP3A to restricted concomitant medications. Table 10 added detailing restricted concomitant medications. CYP3A text is now summarised in Table 10. |
| 5.6.3 Effect of olaparib on other drugs | Sections deleted. Section text is now summarised in Table 10. |
| 5.6.4 Interaction of olaparib and specific co-medications | |
| 5.6.6 Anticoagulant therapy | |
| 5.8.1 Procedures for discontinuation of a patient from study treatment 6.4.4 Reporting of serious adverse events | Reporting of SAEs text amended to specify SAEs, must be reported to AstraZeneca via both the eCRF and paper SAE report to AstraZeneca data entry site (DES) within 24 hours. |
| 6.2.1 Screening procedures | The capturing of adverse events during Screening text has been revised to reflect current practice. |

| | | - | |
|------|----|-----|------|
| Date | 18 | May | 2018 |

| Applicable section number(s)/title | Nature of revision |
|---|---|
| 6.4.3 Recording of adverse events | The recording of adverse events text has been revised to reflect current practice. |
| | A section for recording of adverse events after the 30 day follow up period has been included. |
| | CTCAE grade and changes in CTCAE grade has been included in the list of variables collected for each AE. |
| | New cancers: Text added to say new primary cancers are considered as IDFS event and must also be reported on the endpoint CRF. Patients with new primary cancers which require (neo)adjuvant treatment of any kind for appropriate management must be discontinued from study treatment. |
| | New section for olaparib adverse events of special interest included. These are MDS/AML, new primary malignancy (other than MDS/AML) and pneumonitis. A questionnaire will be sent to any investigator reporting an AESI by AstraZeneca Patient Safety. |
| 6.8 Pharmacokinetics | Text included to clarify samples should be collected preferably on visit 4, day 29, however, samples can also be taken at a later treatment visit, provided that PK consent was obtained beforehand. |
| 11.1.2.1 Overall Survival<br>5.9 Withdrawal from study | Removed survival sweep from the protocol. |
| 12.2.1.1 Primary analysis 12.2.7 Sample size justification | Updated text for the predicted timing for the primary analysis. |
| | Removed text relating to ER+ proportions as the revised predictions are based on the current data which has approximately 15% ER+. |
| 12.2.1.2 Sensitivity analysis | Details of sensitivity analyses included where the results of ER and PgR status from the local and central labs differ in >5% of randomised patients. |
| 12.2.1.3 Subgroup analysis 12.2.2 Analysis of secondary endpoints | Text revised for number of events below which it is not considered appropriate to present analyses. |

| Applicable section number(s)/title | Nature of revision |
|---|---|
| 12.2.3.2 Statistical considerations for patient reported outcomes | Estimates updated based on the sample size increase. |
| 12.2.6 Interim analysis | Updated text for predicted timing for the interim analysis. |
| 12.2.7 Sample size justification | Table 12 Estimated accrual pattern, replaced with new version based on actual accrual pattern between June 2014 and February 2018; now numbered Table 15. Table 13 Estimated annual hazard rates, and text related to this table have been deleted. |
| 13.1 Medical emergencies and contacts | Addresses and roles corrected. |
| 13.2 Overdose | Additional text concerning what constitutes an overdose has been included. |
| 13.3 Pregnancy | Table 16, Pregnancy reporting and handling according to time of diagnosis and Table 17, Reporting outcomes of pregnancy according to time of diagnosis added. |
| 14 List of references | Inclusion of additional references to support new data. |
| Appendix H CYP3A Medications to be avoided with olaparib | Appendix deleted as text now contained within Section 5.6.2 Restricted concomitant medications. |
| Appendix I CPS & EG score | Typographical error in table footnote corrected from 4.1.3a to 4.1.4a. Appendix renumbered to Appendix H. |

Clinical Study Protocol Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5

Date 18 May 2018

#### Version 4, 23 March 2017

Changes to the protocol are summarised below.

- Table of content, the following section is added: 5.5.6.6 Interruptions for intercurrent non-toxicity related events.
- Table of content, List of Appendices is revised due to the new Clinical Study Protocol template:
  - Appendix A Signatures is removed
- Section 4.1 (Inclusion Criteria):

Inclusion criterion 4a

#### **Previous text:**

#### TNBC defined as:

ER and PgR negative defined as IHC nuclear staining <1%. All ER and PgR assessments that are locally available must be negative.

#### Revised text:

#### TNBC defined as:

ER and PgR negative defined as IHC nuclear staining <1%.

#### AND

Inclusion criterion 4b

#### **Previous text:**

#### ER and/or PgR positive, HER2 negative breast cancer defined as:

ER and/or PgR positive defined as IHC nuclear staining ≥1%. Any tumour that has been locally assessed as ER and/or PgR positive in either the core biopsy or the surgical specimen is considered to be ER and/or PgR positive.

#### Revised text:

#### ER and/or PgR positive, HER2 negative breast cancer defined as:

ER and/or PgR positive defined as IHC nuclear staining ≥1%.

The current protocol version incorporated new wording added in the previous amendment which is overly restrictive for patients with tumors classified as triple negative breast cancer based on the receptor status analysis from the core needle biopsy, but who have low levels

of peroxidase staining for ER and PgR in their post-neoadjuvant surgical specimen. By removing the new sentences that allow receptor status to be determined from ANY specimen, we revert to the original protocol version, where the receptor status will be determined from a specimen obtained from treatment naïve tissue. This is supported by the publication describing the CPS+EG score (Mittendorf et al 2011).

• Section 5.5.6.6. (Interruptions for intercurrent non-toxicity related events) is added back in the protocol.

This section was in the original version of the protocol and deleted in error when Amendment 1 was produced. Adding the section back in to the protocol brings it back in line with the guidance in the Investigator Brochure regarding stopping olaparib 3 days prior to planned surgery.

The medical rationale for stopping olaparib 3 days prior to planned surgery is purely a precautionary measure. Three days was chosen based on the half-life of olaparib, to assume that in 3 days most of the drug has been eliminated. There is no data to suggest that olaparib has impact on wound healing, nor have any complications been reported perioperatively related to olaparib.

- Section 13.1 (Medical emergencies and contacts) is updated
- Appendix C (Pharmacogenetics Research) is revised in line with the new Clinical Study Protocol template:
  - Table of contents is removed
  - List of abbreviations and definition of terms is removed
- Appendix D (Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law) is revised in line with the new Clinical Study Protocol template:
  - Title is revised to "Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law"
  - Table of contents is removed
  - The following sentence is added to the Introduction: This Appendix describes the process to be followed in order to identify and appropriately report cases of Hy's Law. It is not intended to be a comprehensive guide to the management of elevated liver biochemistries.
  - Definitions are revised
  - Section 6 "ACTIONS REQUIRED WHEN POTENTIAL HY'S LAWCRITERIA ARE MET BEFORE AND AFTER STARTING STUDY TREATMENT (NOT APPLICABLE)" is removed

Clinical Study Protocol Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5

Date 18 May 2018

#### Version 3, 21 October 2015

Changes to the protocol are summarised below.

Refer to the separate Clinical Study Protocol Amendment document dated 21 October 2015 for the changes made in Revised Clinical Study Protocol Edition 1. Note that the appendices were not updated as part of Revised Clinical Study Protocol Edition 2.

#### Version 2, 14 March 2014

Changes to the protocol are summarised below.

Refer to the separate Clinical Study Protocol Administrative Change document dated 14 March 2014 for the changes made in Revised Clinical Study Protocol Edition 2. Note that the appendices were not updated as part of Revised Clinical Study Protocol Edition 1.

#### Version 1, 25 October 2013

Initial creation

This submission document contains confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

This Clinical Study Protocol has been subject to a peer review according to AstraZeneca Standard procedures. The Clinical Study Protocol is publicly registered and the results are disclosed and/or published according to the AstraZeneca Global Policy on Bioethics and in compliance with prevailing laws and regulations.







## LIST OF OLYMPIA PROTOCOL AUTHORS

| Medical Oncologist, Institute of Cancer Research and King's College London, UK |
|---|
| Medical Oncologist, Alliance, Dana Farber Cancer Institute,<br>USA |
| Medical Oncologist, Sheba Breast Collaborative Group (SBCG), Israel |
| Medical Oncologist, NRG Oncology, Virginia Commonwealth<br>University Massey Cancer Center, USA |
| Research Operations Director, Breast International Group (BIG), Belgium |
| Medical Oncologist, Memorial Sloan-Kettering Cancer<br>Center, USA |
| Study Statistician, NRG Oncology, USA |
| Biostatistics Team Lead, Frontier Science (Scotland) Ltd |
| Medical Research Fellow, Jules Bordet Institute, Belgium |
| Head of Medical Support Team, Jules Bordet Institute,<br>Belgium |
| Medical Oncologist, IBCSG, Hospital of Prato, Italy |
| Medical Oncologist, Perelman School of Medicine, USA |
| Principal Investigator/Senior Biostatistician, Frontier<br>Science and Technology Research Foundation (FSTRF),<br>Boston, MA, USA |
| Medical Oncologist, National Cancer Institute Canada,<br>Clinical Trials Group (NCIC CTG), BC Cancer Agency,<br>Canada |
| Senior Medical Director, Oncology Global Medicines<br>Development, AstraZeneca Gaithersburg, USA |







| Chief Executive Officer, Breast International Group (BIG),<br>Belgium |
|---|
| Surgeon, Austrian Breast and Colorectal Cancer Group<br>(ABCSG), Comprehensive Cancer Center Vienna, Austria |
| Global Product Statistician, AstraZeneca Alderley Park,<br>United Kingdom |
| Managing Director, Frontier Science (Scotland) Ltd |
| Medical Oncologist, Chair, Breast International Group (BIG),<br>Scientific Director, Jules Bordet Institute, Belgium |
| Medical Oncologist, Magee-Womens Hospital of UPMC,<br>NRG Oncology, USA |
| Medical Oncologist, Breast International Group (BIG),<br>Belgium |
| Medical Oncologist, Center for Familial Breast and Ovarian<br>Cancer and Center of Integrated Oncology, Germany |
| Breast Cancer Disease Area Clinical Expert, AstraZeneca<br>Alderley Park, United Kingdom |
| Study Pathologist, Istituto Europeo di Oncologia (IEO),<br>University of Milan, Italy |
| Gynaecologist, German BrEAST Group (GBG), Germany |
| Senior Oncology Research Physician, AstraZeneca Alderley<br>Park, United Kingdom |
| Senior Protocol Statistician, Frontier Science (Scotland) Ltd |
| Senior Protocol Statistician, Frontier Science (Scotland) Ltd |
| Global Product Statistician, AstraZeneca Gaithersburg, USA |
| Medical Director, Breast International Group (BIG),<br>Belgium |
| Global Study Leader, AstraZeneca, Poland |
| Project Manager, Breast International Group (BIG), Belgium |

#### PROTOCOL SYNOPSIS

A randomised, double-blind, parallel group, placebo-controlled multi-centre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy



#### Study centre(s) and number of patients planned

The study will be conducted in approximately 25 countries worldwide. Approximately 700 centres (in the US and Rest of the World countries) will be initiated to randomise approximately 1800 patients. Additional countries and sites may be added dependent on recruitment rates.

Approximately 150 randomised patients\* will be analysed for pharmacokinetic (PK) at those sites that have confirmed that they are able to collect the PK assessment samples. PK sampling will be performed in a subset of patients who sign an optional PK Informed consent.

| Study period | | Phase of development |
|------------------------------------------|---------|----------------------|
| Estimated date of first patient enrolled | Q1 2014 | III |
| Estimated date of last patient completed | 2028 | |

<sup>\*</sup> No placebo samples will be analysed unless requested.

#### **Objectives**

## **Primary Objective**

The primary objective is to assess the effect of adjuvant treatment with olaparib on Invasive Disease Free Survival (IDFS)

## Safety Objective

To assess the safety and tolerability of adjuvant treatment with olaparib

### **Secondary Objectives**

- 1. To assess the effect of adjuvant treatment with olaparib on overall survival (OS)
- 2. To assess the effect of adjuvant treatment with olaparib on Distant Disease Free Survival (DDFS)
- To assess the effect of adjuvant treatment with olaparib on the incidence of new primary contralateral invasive breast cancer, primary contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer
- 4. To assess the effect of olaparib on patient reported outcomes using the FACIT-Fatigue and EORTC QLQ-C30 questionnaires
- 5. To assess the efficacy of olaparib in patients identified as having a deleterious or suspected deleterious variant in either of the *BRCA* genes using variants identified with current and future germline *BRCA* mutation assays (gene sequencing and large rearrangement analysis)
- 6. To determine the exposure to olaparib (in plasma) in patients receiving olaparib as adjuvant therapy





#### Study delivery model

This is a collaborative study being coordinated worldwide by the Breast International Group (BIG) in partnership with Frontier Science (FS), NRG Oncology (NCI supported National Clinical Trials Network Group) and AstraZeneca (AZ). Two versions of this protocol have been written to cover this global adjuvant breast cancer study. One protocol version covers all patients recruited outside of the US (where AZ is the sponsor) and one protocol version covers patients recruited within the US (where NRG Oncology is the sponsor). The two versions of the protocol are identical in terms of study objectives and scientific content and only differ in logistical content appropriate for the country(ies) they cover (i.e. drug distribution, mechanisms for SAE reporting during the study, etc). Based on current recruitment rates, it is expected that approximately 230 patients will be randomised under the US protocol and approximately 1570 will be randomised under the Rest of the World protocol.

The trial will use one randomisation system and report as one single study. The initial collection of the patients' data will be done using two databases (one for the US patients and one for all other patients outside of the US). The two databases will be set up using the same standards and eCRFs to ensure consistency in the data collection. The data from both databases will be combined into a single consolidated database at regular, pre-specified intervals. All study endpoints as well as reports for periodic review by the Independent Data Monitoring Committee (IDMC) will be analysed and reported from the single combined reporting database, held by Frontier Science on behalf of BIG.

#### Study design

This is a randomised, double-blind, parallel group, placebo-controlled multi-centre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy.

Patients will be randomised in a 1:1 ratio to either olaparib or placebo. Randomisation will be stratified by hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC), by prior neoadjuvant versus adjuvant chemotherapy, and prior platinum use for breast cancer (yes versus no).

Eligible patients with deleterious or suspected deleterious gBRCA mutations and high risk HER2 negative breast cancer should be randomised in the trial ideally within a maximum of 8 weeks of completing their last treatment modality (chemotherapy and definitive local or locoregional treatment), but in no case longer than 12 weeks. Randomised patients will receive study treatment for up to a maximum of 12 months. All patients will have safety assessments every 2 weeks during the first month, every 4 weeks for the following 5 months (up to week 24) and 3 monthly for the remaining 6 months of study treatment plus 30 days after its discontinuation. All randomised patients will have clinical assessment visits for approximately 10 years following their randomisation into the study, or until an IDFS endpoint due to a breast cancer related distant relapse, whichever comes first. They then enter the annual survival follow-up phase of the trial, which will continue until 10 years after the last patient is randomised. No clinic visits will be required during the survival follow-up phase; information may be collected via telephone, medical records or death registries.

#### Target patient population

Patients eligible for the trial are those with a deleterious or suspected deleterious germline *BRCA* mutation (defined by local or central Myriad testing) with high risk HER2 negative primary breast cancer who have completed definitive local treatment, and neoadjuvant or adjuvant chemotherapy. Definitions of high risk HER2 negative patients are provided below.

- 1. For patients who underwent initial surgery and received adjuvant chemotherapy
  - TNBC patients must have been axillary node-positive (≥pN1, any tumour size) or axillary node negative (pN0) with invasive primary tumour pathological size > 2 cm (≥pT2)
  - ER and/or PgR positive/HER2 negative patients must have had ≥4 pathologically confirmed positive lymph nodes.
- 2. For patients who underwent neoadjuvant chemotherapy followed by surgery
  - TNBC patients must have residual invasive breast cancer in the breast and/or resected lymph nodes (non pCR)
  - ER and/or PgR positive/HER 2 negative patients must have residual invasive cancer in the breast and/or the resected lymph nodes (non pCR) AND a CPS&EG score ≥3 (Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS)- a disease scoring system). Instructions how to calculate CPS&EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix H.

#### Germline BRCA1 and BRCA2 (gBRCA) testing

Local gBRCA testing results, if available, can be used for establishing eligibility. If local gBRCA testing results are not available, central testing will be provided for those patients who otherwise appear to be eligible. Irrespective of the availability of local gBRCA testing results, all patients must provide a sample for central gBRCA testing.

# Central tumour analyses (e.g. somatic *BRCA1/2* functional status, ER/PgR and HER2 status)

Archival tumour samples must be provided for all patients.

For adjuvant patients, this refers to the surgical specimen; for neoadjuvant patients, both the pre-treatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and reembedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required.

## Study treatment, dosage and mode of administration

AstraZeneca's Pharmaceutical Development, R&D Supply Chain will supply olaparib and matching placebo to the investigator as green film-coated tablets.

Patients will be randomised in a 1:1 ratio to one of the following treatments:

- 12 months treatment with olaparib tablets p.o. 300 mg twice daily (two 150 mg tablets in the morning and two 150 mg tablets in the evening)
- 12 months treatment with matching placebo tablets p.o. twice daily (two tablets in the morning and two tablets in the evening)

#### Stratification

Patients will be stratified at randomisation by the following baseline factors:

- Hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC)
  - NOTE: In cases of multifocal, multicentric or synchronous bilateral invasive disease, stratification is based on the status of the lesion considered at highest risk (at the investigator's discretion) that was used to determine eligibility.
- Neoadjuvant versus adjuvant chemotherapy
- Platinum therapy for current breast cancer: Yes/No

Within this study, patients will not be provided with olaparib post discontinuation of study treatment. Patients and investigators will not be routinely unblinded to study treatment prior to the final overall survival (OS) analysis. Unblinding is allowed only in case of compelling medical or safety reasons (Section 5.4.2).

#### Outcome(s):

- Primary outcome
  - Invasive Disease Free Survival (IDFS)
- Secondary outcomes
  - Overall Survival (OS)
  - Distant Disease Free Survival (DDFS)
  - New primary contralateral breast cancers (invasive and non-invasive), new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancers in patients at risk for these events

- FACIT-Fatigue symptom scale score and EORTC-QLQ-C30 global health status, functional, and symptoms scales/items scores
- IDFS, DDFS and OS based on patients with gBRCA mutations confirmed by the central test (only required if population differs from the ITT (intention to treat) population)
- Pharmacokinetic analysis
- Safety outcomes
  - Adverse Events (AE), physical examination, vital signs including blood pressure (BP), pulse, and laboratory findings including clinical chemistry and haematology



#### Statistical methods

The primary endpoint of the study is IDFS and patients will be randomised 1:1 to either olaparib 300 mg b.i.d. (twice daily) or matching placebo.

Approximately 1800 patients will be randomised into the study. If the true hazard ratio for the comparison of olaparib versus placebo in terms of IDFS is 0.7 then with 330 events, the analysis of IDFS will have 90% power to demonstrate a statistically significant difference in IDFS, assuming a 2-sided 5% significance level. It is estimated the study will take approximately 5 years to complete recruitment of 1800 patients. The primary analysis will be triggered by the occurrence of 330 IDFS events (required for overall 90% power to detect a HR of 0.7). Assuming a non-uniform recruitment, the primary analysis is estimated to occur approximately 6 years from the start of randomisation.

An interim analysis for superiority will be performed once a minimum of 165 IDFS events have been observed from the first 900 patients recruited. It is estimated that this analysis will occur approximately 5.3 years after the first patient is randomised. Consideration of futility will also be made at the time of interim analysis.

Safety data will be summarised descriptively in terms of AEs, vital signs, clinical chemistry & haematology and physical exam and will include all patients who received at least one dose of olaparib or placebo.

Patient reported outcomes and health related quality of life (HRQoL) will be assessed through the planned correlative study using the FACIT-Fatigue and the EORTC QLQ-C30 questionnaires.

An analysis of IDFS, DDFS and OS will be conducted based on patients with gBRCA mutations confirmed by the central test, if this population differs from the primary ITT population. Similar sensitivity analyses will be performed based on ER and/or PgR positive/HER2 negative and TNBC subsets as defined by the central laboratory testing.

Full details of all the statistical analyses will be documented in the SAP. Version 1.0 of the SAP will be prepared prior to first subject in (FSI).

#### Pharmacokinetic analysis

The plasma concentration-time data will be analysed by non-linear mixed effects modelling in order to evaluate the pharmacokinetic characteristics of olaparib, quantify variability in the pharmacokinetics, identify demographic or pathophysiological covariates, which may explain the observed variability and explore exposure-response relationships.

TABLE OF CONTENTS

#### TITLE PAGE......1 VERSION HISTORY \_\_\_\_\_\_2 LIST OF ABBREVIATIONS AND DEFINITION OF TERMS.......28 1. Background 33 1.1 1.1.1 Breast cancer and its treatment 33 1.1.2 1.1.3 Adjuvant chemotherapy for TNBC......34 1.1.4 Neoadjuvant chemotherapy for TNBC .......34 1.1.5 ER/PgR positive HER2 negative breast cancer with germline BRCA 116 PARP inhibition as a therapeutic strategy target for *BRCA* mutated breast cancer 36 1.1.7 Pre-clinical experience 36 1.1.8 1.1.9 1.1.9.1 1.2 1.3 1.3.1 1.4 Benefit/risk and ethical assessment 41 STUDY OBJECTIVES......46 2. 2.1 2.2 Secondary objectives 46 2.3 ......46 3. 3.1 3.2

**PAGE** 

| 3.2.1 | Rationale for study design | 62 |
|---|---|---|
| 3.2.2 | Rationale for patient reported outcomes | |
| 3.2.3 | Study Population | 64 |
| 4. | PATIENT SELECTION CRITERIA | 65 |
| 4.1 | Inclusion criteria | 65 |
| 4.2 | Exclusion criteria | 70 |
| 5. | STUDY CONDUCT | 72 |
| 5.1<br>5.1.1<br>5.1.2 | Restrictions during the study Meals and dietary restrictions Contraception | 72 |
| 5.2<br>5.2.1 | Patient enrolment and randomisation and initiation of study treatment | |
| 5.3 | Procedures for handling patients incorrectly enrolled or randomised or initiated on study treatment | 74 |
| 5.4 | Blinding and procedures for unblinding the study | |
| 5.4.1<br>5.4.2 | Methods for ensuring blinding | |
| 5.5 | Treatments | |
| 5.5.1 | Identity of study treatment | |
| 5.5.2 | Doses and treatment regimens | |
| 5.5.2.1 | Olaparib and matching placebo (study treatment) | |
| 5.5.3 | Additional study drug - Not applicable | |
| 5.5.4<br>5.5.5 | LabellingStorage | |
| 5.5.6 | Management of toxicity of study treatment | |
| 5.5.6.1 | Study therapy following breast cancer recurrence or second primary cancer | |
| 5.5.6.2 | Olaparib/placebo dose levels | |
| 5.5.6.3 | Renal impairment | |
| 5.5.6.4 | Management of haematological toxicity | |
| 5.5.6.5 | Management of new or worsening pulmonary symptoms | |
| 5.5.6.6 | Management of nausea and vomiting | |
| 5.5.6.7 | Interruptions for intercurrent non-toxicity related events | 83 |
| 5.6 | Concomitant and subsequent treatment(s) | |
| 5.6.1 | Administration of endocrine therapy | |
| 5.6.2 | Restricted concomitant medications | |
| 5.6.3 | Anti-emetics/Anti-diarrheals | |
| 5.6.4 | Live virus and bacterial vaccines. | |
| 5.7 | Treatment compliance | |
| 5.7.1 | Accountability | 87 |

| 5.8 | Discontinuation of study treatment | 87 |
|---|---|---|
| 5.8.1 | Procedures for discontinuation of a patient from study treatment | 88 |
| 5.9 | Withdrawal from study | 89 |
| 6. | COLLECTION OF STUDY VARIABLES | 90 |
| 6.1 | Recording of data | 90 |
| 6.2 | Study procedures | 90 |
| 6.2.1 | Screening procedures | |
| 6.2.2 | On-treatment assessments | |
| 6.2.3 | Efficacy follow-up assessments | 95 |
| 6.2.4 | Safety follow-up assessments 30 days after last dose of olaparib/placebo | 95 |
| 6.2.5 | Patient management post-primary analysis | 96 |
| 6.2.6 | Patient management post-final analysis | 96 |
| 6.3 | Efficacy | 96 |
| 6.3.1 | Tumour evaluation | |
| 6.4 | Safety | 98 |
| 6.4.1 | Definition of adverse event (AE) | 98 |
| 6.4.2 | Definitions of serious adverse event (SAE) | |
| 6.4.3 | Recording of adverse events | 99 |
| 6.4.4 | Reporting of serious adverse events | |
| 6.4.5 | Laboratory safety assessment | |
| 6.4.5.1 | Full haematology assessments for safety | |
| 6.4.5.2 | Coagulation | |
| 6.4.5.3 | Clinical chemistry assessments for safety | |
| 6.4.5.4 | Urinalysis | |
| 6.4.5.5 | Bone marrow or blood cytogenetic samples | |
| 6.4.6 | Physical examination | |
| 6.4.7 | ECG | |
| 6.4.7.1 | Resting 12-lead ECG | |
| 6.4.8 | Vital signs | |
| 6.4.8.1 | Pulse and blood pressure | |
| 6.4.8.2 | Body temperature | |
| 6.4.9 | Other safety assessments | |
| 6.4.9.1 | Serum or urine pregnancy test | 107 |
| 6.5 | Patient reported outcomes (PRO) | 108 |
| 6.5.1 | FACIT-Fatigue | 108 |
| 6.5.2 | EORTC QLQ-C30 | |
| 6.5.3 | Administration of PRO questionnaires | 109 |
| 6.6 | Biomarkers | |
| 6.6.1 | Biomarker samples | 110 |
| 6.6.2 | Collection of blood sample for Myriad germline BRCA1 and BRCA2 | |
| | testing | 111 |

| 6.6.2.1 | Collection of a blood sample for assessment of current and future <i>BRCA</i> mutation assay(s) | | |
|---|---|---|---|
| | mutation assay(s) | 11 | . 4 |
| g. | | | |
| 5.0 | | orace | 1 101 |
| | | 11 | |
| 6.8 | <del>.</del> | | |
| 6.8.1 | Pharmacokinetics (optional) | | |
| 6.8.2 | Collection of samples | 11 | 14 |
| 6.8.3 | Determination of drug concentration | 11 | 15 |
| 6.9 | Health economics | | |
| 6.9.1 | Resource use (serious adverse events) | | |
| 7. | BIOLOGICAL SAMPLING PROCEDURES | | |
| 7.1 | Volume of blood | 11 | 15 |
| 7.2 | Handling, storage and destruction of biological samples | | |
| 7.2.2 | Pharmacokinetic samples | 11<br>11 | 17 |
| 7.3 | Labeling and shipment of biohazard samples | 11 | 18 |
| 7.4 | Chain of custody of biological samples | 11 | 18 |
| 7.5 | Withdrawal of informed consent for donated biological samples. | 11 | 18 |
| 8. | ETHICAL AND REGULATORY REQUIREMENTS | 12 | 20 |
| 8.1 | Ethical conduct of the study | 12 | 20 |
| 8.2 | Patient data protection | 12 | 20 |
| 8.3 | Ethics and regulatory review | 12 | 20 |
| 8.4 | Informed consent | 12 | 21 |
| 8.5 | Changes to the protocol and informed consent form | 12 | 22 |
| 8.6 | Audits and inspections | 12 | 22 |
| 9. | STUDY MANAGEMENT | 12 | 22 |
| 9.1 | Pre-study activities | 12 | 22 |
| 9.2 | Training of study site personnel | 12 | 23 |

| Monitoring of the study | |
|---|---|
| Study agreements Archiving of study documents | |
| Study timetable and end of study | 124 |
| DATA MANAGEMENT | . 124 |
| EVALUATION AND CALCULATION OF VARIABLES | . 125 |
| Calculation or derivation of efficacy variable(s) | 125 |
| • 1 | |
| Distant disease free survival (DDFS) | |
| Incidence of contralateral invasive breast cancer, contralateral non-<br>invasive breast cancer, new primary ovarian cancer, new primary fallopian<br>tube cancer and new primary peritoneal cancer | 128 |
| Calculation or derivation of safety variable(s) Other significant adverse events (OAE) | |
| Calculation or derivation of patient reported outcome variables | 129 |
| Calculation or derivation of pharmacokinetic variables | . 129 |
| Calculation or derivation of pharmacodynamic variable(s) - not applicable | . 129 |
| Calculation or derivation of variables | . 129 |
| Calculation or derivation of health economic variables –not applicable | 129 |
| STATISTICAL METHODS AND SAMPLE SIZE DETERMINATION | 129 |
| Description of analysis sets Full analysis set Safety analysis set PK analysis set | 129<br>130 |
| Analysis of primary endpoint | 131 |
| Analysis of Interaction | |
| Analysis of secondary endpoints | |
| Analysis of patient reported outcomes | |
| 1 1 | |
| | Source data Study agreements |

| | | 139 |
|---|---|---|
| 12.2.5 | Multiplicity strategy for primary and key secondary endpoints | 140 |
| 12.2.6<br>12.2.7 | Interim analysis | |
| 12.3 | Independent Data monitoring committee | |
| 13. | IMPORTANT MEDICAL PROCEDURES TO BE FOLLOWED BY THE | 1 10 |
| 13. | INVESTIGATOR | 147 |
| 13.1 | Medical emergencies and contacts. | 147 |
| 13.2 | Overdose | 148 |
| 13.3 | Pregnancy | |
| 13.3.1<br>13.3.2 | Maternal exposure Paternal exposure | |
| 14. | LIST OF REFERENCES | |
| LIST O | F TABLES | |
| Table 1 | Study Schedule - Screening (PART 1 and PART 2) | 52 |
| Table 2 | Study Schedule – On treatment (Year 1) | 55 |
| Table 3 | Study Schedule - Follow-up Visits (Year 2 onwards) | 59 |
| Table 4 | Identity of study treatment | 76 |
| Table 5 | Study treatment doses and treatment regimens | 77 |
| Table 6 | Olaparib/placebo dose levels | 79 |
| Table 7 | Mandatory Treatment for Hematologic Toxicity and Treatment Guidance for other olaparib/placebo Toxicities | 80 |
| Table 8 | Dose reduction for study treatment to manage moderate renal impairment | 81 |
| Table 9 | Dose reduction for study treatment with concurrent use of a strong or moderate CYP3A inhibitor | 82 |
| Table 10 | Restricted concomitant medications | 85 |
| Table 11 | Samples for Biomarker Research | 110 |
| Table 12 | Volume of blood to be drawn from each patient | 116 |
| Table 13 | Summary of Outcome Variables and Analysis Populations | 130 |
| Table 14 | Summary of 2-sided significance levels and total alpha spend across the endpoints and analyses | 143 |
| Table 15 | Actual accrual between June 2014 and February 2018 | 145 |

| Table 16 | Pregnancy reporting and handling according to time of diagnosis | 149 |
|---|---|---|
| Table 17 | Reporting outcomes of pregnancy according to time of diagnosis | 150 |
| Table 18 | Point assignments for the CPS + EG staging system | 176 |
| LIST OF FIG | GURES | |
| Figure 1 | Study Flow Chart | 50 |
| Figure 2 | Screening Plan | 51 |
| Figure 3 | Multiple testing procedure | 141 |
| LIST OF AP | PENDICES | |
| Appendix A | Additional Safety Information | 159 |
| Appendix B | International Airline Transportation Association (IATA) 6.2 Guidance Document | 161 |
| | | 162 |
| Appendix D | Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law | 166 |
| Appendix E | Acceptable Birth Control Methods | 170 |
| Appendix F | ECOG Performance Status | 172 |
| Appendix G | Patient Reported Outcomes (FACIT-Fatigue, EORTC QLQ-C30) | 173 |
| Appendix H | CPS & EG score. | 176 |

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

The following abbreviations and special terms are used in this study Clinical Study Protocol.

| Abbreviation or special term | Explanation |
|---|---|
| AE | Adverse event (see definition in Section 6.4.1) |
| AESI | Adverse event of special interest |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AML | Acute Myeloid Leukaemia |
| ANC | Absolute neutrophil count |
| APTT | Activated Partial Thromboblastin Time |
| ASCO | American Society of Clinical Oncology |
| AST | Aspartate aminotransferase |
| AUC | Area Under Curve |
| b.i.d. | Twice daily |
| BP | Blood Pressure |
| BRCA | Breast cancer susceptibility gene |
| BUN | Blood Urea Nitrogen |
| CA-125 | Cancer antigen-125 |
| CfDNA | Circulating free DNA |
| СНО | Chinese hamster ovary |
| CI | Confidence Interval |
| Cmax <sub>ss</sub> | Maximum concentration at steady state |
| Cmin <sub>ss</sub> | Minimum concentration at steady state |
| CNS | Central Nervous System |
| CPS&EG | Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS)- a disease scoring system |
| CR | Complete Response |
| CRF (eCRF) | Case Report Form (electronic/paper) |
| CRO | Contract Research Organisation |
| CSA | Clinical Study Agreement |
| CSR | Clinical Study Report |
| CT | Computerised Tomography |

| Abbreviation or special term | Explanation |
|---|---|
| CTCAE | Common Terminology Criteria for Adverse Event |
| DAE | Discontinuation of study treatment due to Adverse Event |
| DCIS | Ductal carcinoma in situ |
| DCO | Data cut off |
| DDFS | Distant disease free survival |
| DES | Data entry site |
| DFS | Disease free survival |
| DNA | Deoxyribonucleic acid |
| DSB | Double strand break |
| DUS | Disease under Study |
| EC | Ethics Committee, synonymous to Institutional Review Board (IRB) and Independent Ethics Committee (IEC) |
| ECG | Electrocardiogram |
| ECOG performance status | Eastern Cooperative Oncology Group performance status using scales and criteria to assess how a patient's disease is progressing |
| EORTC QLQ-C30 | The European Organisation for Research and Treatment of Cancer -Quality of Life Questionnaire-Core questions 30 |
| ER | Estrogen receptor |
| ESMO | European Society for Medical Oncology |
| ESTRO | European Society for Radiation and Oncology |
| FACIT-Fatigue | Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue<br>Measurement questionnaire |
| FAS | Full Analysis Set |
| FFPE | Formalin Fixed Paraffin Embedded |
| FSH | Follicle Stimulating Hormone |
| gBRCA mutation or gBRCAm | The term "gBRCA mutation" is used to refer to a germline BRCA1 or BRCA2 mutation classified as "deleterious" or "suspected deleterious" in accordance with the American College of Medical Genetics and Genomics recommendations for standards for interpretation and reporting of sequence variants |
| GCP | Good Clinical Practice |
| G-CSF | Granulocyte Colony Stimulating Factor |
| GMP | Good Manufacturing Practice |
| Hgb | Hemoglobin |

| Abbreviation or special term | Explanation |
|---|---|
| HDPE | High Density Polyethylene |
| HER2 | Human Epidermal Growth Factor Receptor 2 |
| HR | Hazard Ratio |
| HRD | Homologous Recombination Deficiency |
| HRQoL | Health Related Quality of Life |
| IB | Investigators Brochure |
| ICH | International Conference on Harmonisation |
| International<br>Co-ordinating<br>investigator | If a study is conducted in several countries the International Co-ordinating Investigator is the Investigator co-ordinating the investigators and/or activities internationally. |
| IDFS | Invasive Disease-free Survival |
| IDMC | Independent Data Monitoring Committee |
| IHC | Immunohistochemistry |
| IIBTR | Ipsilateral invasive breast tumour recurrence |
| INR | International Normalised Ratio |
| IPCW | Inverse Probability of Censoring Weighting |
| ISH | In Situ Hybridisation (includes FISH, DISH, CISH) |
| ISS | Investigator Sponsored Study |
| ITT | Intention To Treat |
| IVRS | Interactive Voice Response System |
| IWRS | Interactive Web Response System |
| KM | Kaplan-Meier |
| LDH | Lactic Dehydrogenase |
| LIMS | Laboratory Information Management System |
| LLOQ | Lower Limit of Quantification |
| LSI | Last Subject in |
| LSLV | Last Subject Last Visit |
| MCH | Mean Cell Haemoglobin |
| MCHC | Mean Cell Haemoglobin Concentration |
| MCV | Mean Cell Volume |
| MDS | Myelodysplastic Syndrome |
| MMRM | Mixed Model for Repeated Measures |

| Abbreviation or special term | Explanation |
|---|---|
| MRI | Magnetic Resonance Image |
| MTD | Maximum Tolerated Dose |
| MTP | Multiple testing procedure |
| NCCN | National Comprehensive Cancer Network |
| NSABP | National Surgical Adjuvant Breast and Bowel Project |
| NSCLC | None Small cell lung cancer |
| OAE | Other Significant Adverse Event (see definition in Section 11.2.1) |
| OD | Once Daily |
| OR | Objective Response |
| ORR | Objective Response Rate |
| OS | Overall survival |
| PARP | Polyadenosine 5'diphosphoribase [poly (ADP ribose)] polymerisation |
| pCR | Pathological Complete Response |
| PD | Pharmacodynamics |
| PFS | Progression Free Survival |
| PFS2 | Time to second progression |
| PgR | Progesterone receptor |
| PGx | Pharmacogenetic research |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| PO | Per Os (by mouth) |
| PRO | Patient Reported Outcome |
| QOL | Quality of Life |
| QT/QTc | A measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (c indicates the corrected value for this time period) |
| RBC | Red Blood Cells |
| RECIST | Response Evaluation Criteira in Solid tumours. This study will use modified RECIST version 1.1. |
| REML | Restricted Maximum Likelihood |
| RPSFT | Rank Preserving Structural Failure Time |
| SAE | Serious adverse event (see definition in Section 6.4.2). |

| Abbreviation or special term | Explanation |
|---|---|
| SAP | Statistical Analysis Plan |
| SCLC | Small Cell Lung Cancer |
| SD | Stable Disease |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic-pyruvic transaminase |
| SNB | Sentinel Node Biopsy |
| SSB | Single Strand Break |
| STEEP | Standardised Terms for Efficacy Endpoints |
| Study treatment | Study treatment is the treatment to which patient was randomised. In this study it is either olaparib or placebo |
| TN1-3 | TNM classification. Axillary node positive disease regardless of the tumour size |
| TNBC | Triple negative breast cancer |
| TPC | Chemotherapy of physician's choice |
| ULN | Upper Limit of Normal |
| WBC | White Blood Cells |
| WBDC | Web Based Data Capture |
| Wt | Wildtype (patients without evidence of <i>BRCA1</i> or <i>BRCA2</i> deleterious or suspected deleterious mutations) |

#### 1. INTRODUCTION

## 1.1 Background

#### 1.1.1 Breast cancer and its treatment

Breast cancer is a life-threatening disease and is the second leading cause of cancer death among women. In 2013, an estimated 232,340 new cases of invasive breast cancer were expected to be diagnosed among US women, and approximately 39,620 women were expected to die from breast cancer (American Cancer Society 2013). In the European Community, the estimated age adjusted annual incidence in 2008 was 88.4/100 000 and the mortality 24.3/100 000 (Aebi et al 2011).

Approximately 5% of breast cancers are associated with a mutation in the *BRCA1* and/or *BRCA2* gene with approximately 3% associated with the *BRCA1* gene (generally presenting with TNBC phenotype) and approximately 2% associated with the *BRCA2* gene (generally ER/PgR positive phenotype). In the general population, *BRCA* mutation carriers have an increased relative risk of breast cancer. The presence of *BRCA1* mutations is associated with a lifetime risk of breast cancer of 60 to 70% and a lifetime risk of ovarian cancer of 20 to 45% (Antoniou et al 2003). *BRCA2* mutations are associated with lifetime risk of breast cancer of 40 to 60% in women and 5 to 10% in men and a lifetime risk of ovarian cancer of 10 to 20%. Rare individuals carry deleterious mutations in both *BRCA1* and *BRCA2* genes.

In breast cancer, there are differences between *BRCA1* and *BRCA2* mutation carriers. Approximately 70% of breast cancer patients with *BRCA1* mutations present as triple negative breast cancer (TNBC). In contrast, patients carrying mutations in the *BRCA2* gene are more likely to be positive for expression of the estrogen receptor in their breast cancer while approximately 20% will have triple negative cancers (Mavaddat et al 2012).

Although there are phenotypic differences in breast cancers resulting from *BRCA1* or *BRCA2* mutations, their important commonality is that mutations in either gene result in tumours that are deficient in homologous recombination, making both appropriate for treatment with polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerisation (PARP) inhibitors whereby the process of synthetic lethality can be exploited. In a previous AstraZeneca sponsored Phase II proof of concept study in patients with breast cancer carrying *BRCA* mutations (Study D0810C00008), approximately 60% of cases were *BRCA1* mutations (the other 40% were *BRCA2* mutations) with 55% of tumours overall triple negative in phenotype. In this study, anti-tumour activity was seen in patients with either *BRCA1* or *BRCA2* mutations (Tutt et al 2010).

Given the small size of the *BRCA* subpopulation in breast cancer, information comparing the outcome from this subpopulation with the overall breast cancer population is based on reports from a number of small studies (Robson et al 2004, Rennert et al 2007, Bordeleau et al 2011, Goodwin et al 2012), and firm conclusions cannot be drawn. The overall body of evidence suggests that once baseline prognostic factors (such as hormone receptor and HER2 status) and treatment are taken into account, patients with *BRCA* mutations have a similar outcome to

their sporadic counterparts (Huzarski et al 2013). This is in contrast to patients with *BRCA1/BRCA2*-related ovarian cancer who have an improved survival compared with non-carriers, particularly if they receive platinum-based therapy.

Currently, there are no approved treatments specific for germline *BRCA*1/2 mutated breast cancer patients and these patients are treated according to their hormone receptor and HER2 status.

#### 1.1.2 Triple Negative Breast Cancer (TNBC)

TNBC is a particular subset of breast cancer defined by lack or low immunohistochemical expression of ER, PgR and HER2 (IHC 0, 1+ or 2+ /FISH non-amplified) and represents approximately 12-17% of breast cancers overall (Foulkes et al 2010). Although it is a heterogeneous group, patients with TNBC have generally poor prognosis (Metzger-Filho et al 2010). The fundamental clinical characteristic of TNBC is early recurrence with likely early visceral metastases, as well as shorter period from time to recurrence to death as compared with other breast cancer types (Dent et al 2007). Chemotherapy remains the ultimate treatment option for those patients with varied impact on long-term prognosis. No targeted treatment has been developed for TNBC, in contrast to endocrine treatment and anti-HER2 treatments, which have significantly improved the clinical outcomes in ER/PgR positive and HER2 positive breast cancer patients, respectively. The standard clinical practice for early stage TNBC following completion of definitive local and systemic chemotherapy treatment is observation. Therefore, TNBC patients having a poor prognosis and limited treatment options present an unmet need for targeted treatment development.

#### 1.1.3 Adjuvant chemotherapy for TNBC

The majority of patients presenting with early TNBC receive adjuvant chemotherapy. The first randomised Phase III study specifically conducted in early TNBC is the BEATRICE study- an Open Label 2-arm Study to Evaluate the Impact of Adjuvant Bevacizumab on Invasive Disease Free Survival in Triple Negative Breast Cancer (Cameron et al 2013). In this study, 2591 patients with resected early TNBC were randomised to receive adjuvant anthracycline and/or taxane chemotherapy with or without bevacizumab, followed by bevacizumab monotherapy for 12 months. The trial did not meet its primary objective of prolonging invasive disease free survival (IDFS). The 3-year IDFS for both arms of the study was approximately 83%. It was commented that this 3-year IDFS was better than anticipated; however, it should be noted that 63% of patients in the trial were node negative, and ~36% had tumours < 2cm. There are no published robust long-term data for subgroups (e.g. different nodal status or *BRCA* mutated tumours) of TNBC treated with standard of care chemotherapy.

#### 1.1.4 Neoadjuvant chemotherapy for TNBC

It is assumed that approximately a third to half of the patients with TNBC will receive chemotherapy in the neoadjuvant setting. The key prognostic information following neoadjuvant chemotherapy is whether patients have residual disease or have had a pathological complete response (pCR; absence of any residual invasive cancer on hematoxylin

and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes). Individual patients who achieve pCR following neoadjuvant chemotherapy have significant improvement in both disease-free survival (hazard ratio (HR) 0.48, 95% CI: 0.37-0.63) and overall survival (HR 0.48, 95% CI: 0.33-0.69) compared with patients with residual invasive disease (Mieog et al 2007). An M.D. Anderson, single institution experience reported 46% pCR rate achieved in a small number of BRCA1 mutated (n=57) breast cancer patients following anthracycline/taxane neoadjuvant chemotherapy (Arun et al 2011). In TNBC, the prognosis of patients who experience pCR is very similar to that for patients with other breast cancer subtypes with less than 10% developing a distant recurrence at 5 years. However, those patients with TNBC who do not experience pCR have a much poorer prognosis (Liedtke et al 2008, Carey 2011). A recently published meta-analysis of anthracycline and taxane containing neoadjuvant chemotherapy trials showed that of 911 patients with TNBC, 282 patients (31%) experienced a pCR (Von Minckwitz et al 2012). Compared with these patients, patients who did not experience a pCR were at higher risk of earlier recurrence over time (HR 6.02, 95% CI: 3.92-9.25) and at higher risk of earlier death over time (HR 12.41, 95% CI: 5.82-26.49). These results highlight the need to develop further treatment options to improve the prognosis of TNBC patients who do not achieve pCR after neoadjuvant chemotherapy.

## 1.1.5 ER/PgR positive HER2 negative breast cancer with germline *BRCA* mutations

While most breast cancers arising in patients with germline *BRCA* mutations are associated histologically with the TNBC phenotype, some - particularly those with underlying germline *BRCA*2 mutations - display a non-TNBC phenotype (Honrado et al 2006; Mavaddat et al 2012). Atchley et al 2008 found positivity for ER/PgR receptor expression in more than 60% of patients with documented germline *BRCA*2 mutations and in about 30% of patients with documented *BRCA*1 mutations.

Traditionally, these patients have been treated in the same manner as ER/PgR positive patients with either unknown or wildtype *BRCA* status. However, ER/PgR positive, HER2 negative patients with *BRCA2* mutations have been shown to have higher risk of recurrence and death than similar patients without mutations (Tryggvadottir et al 2013), suggesting that the current management of these patients could be suboptimal.

This could be particularly true for high-risk ER/PgR positive, HER2 negative breast cancer patients. Results from NSABP B-38, a trial which employed modern anthracycline and taxane regimens in the adjuvant setting, showed that hormone receptor positive patients with 4 or more positive axillary nodes at surgery had a 3 year DFS of 83%, which is comparable to the 3-year DFS of node negative TNBC (Swain et al 2013).

Similar considerations can be applied to the neoadjuvant setting. In a recently published, FDA co-sponsored meta-analysis looking into the association between the achievement of pCR and long-term clinical benefit, pCR rates in patients with ER and/or PgR positive, HER2 negative tumours were between 8% to 16%, as opposed to 34% in TNBC (Cortazar et al 2014). While all published subgroups in that analysis indicated clinical benefit (longer recurrence-free survival) for those patients achieving a pCR, the associated prognostic value varied

quantitatively as evidenced by HRs between 0.24 (TNBC patients) and 0.63 (low grade ER and/or PgR positive, HER2 negative tumours with an upper bound of the confidence interval [CI] being slightly above 1.0). A robust association between failure to achieve pCR and event-free survival was demonstrated in patients with ER and/or PgR positive, HER2 negative Grade 3 tumours. Specifically, the HR for event-free survival in that patient group was found to be almost the same (0.27) as the HR for event-free survival in patients with TNBC (0.24). This demonstrates that for carefully selected, high risk ER and/or PgR positive, HER2 negative patients, failure to achieve pCR can have relatively similar prognostic value as in patients with TNBC who have residual disease after neoadjuvant chemotherapy.

## 1.1.6 PARP inhibition as a therapeutic strategy target for *BRCA* mutated breast cancer

PARP inhibition is a novel approach to targeting tumours with deficiencies in DNA repair mechanisms. PARP enzymes are essential for repairing DNA single strand breaks (SSBs). Inhibiting PARPs leads to the persistence of SSBs, which are then converted to the more serious DNA double strand breaks (DSBs) during the process of DNA replication. During the process of cell division, DSBs can be efficiently repaired in normal cells by homologous recombination repair. Tumours with homologous recombination deficiencies (HRD), such as ovarian or breast cancers in patients with germline *BRCA1/2* mutations, cannot accurately repair the DNA damage, which may become lethal to cells as it accumulates. In such tumour types, olaparib may offer a potentially efficacious and less toxic cancer treatment compared with currently available chemotherapy regimens.

BRCA1 and BRCA2 defective tumours are intrinsically sensitive to PARP inhibitors, both in tumour models *in vivo* (Rottenberg et al 2008, Hay et al 2009) and in the clinic (Fong et al 2009). The mechanism of action for olaparib results from the trapping of inactive PARP onto the single-strand breaks preventing their repair (Helleday 2011, Murai et al 2012). Persistence of SSBs during DNA replication results in their conversion into the more serious DNA DSBs that would normally be repaired by homologous recombination repair. Olaparib has been shown to inhibit selected tumour cell lines in vitro and in xenograft and primary explant models as well as in genetic BRCA knockout models, either as a stand-alone treatment or in combination with established chemotherapies (data on file at AstraZeneca).

Olaparib is a potent PARP inhibitor (PARP-1, -2 and -3) that is being developed as an oral therapy, both as a monotherapy (including maintenance) and for combination with chemotherapy and other anti-cancer agents.

#### 1.1.7 Pre-clinical experience

The pre-clinical experience is fully described in the current version of the olaparib IB.

## 1.1.8 Toxicology and safety pharmacology summary

Olaparib has been tested in a standard range of safety pharmacology studies e.g., dog cardiovascular and respiratory function tests, and the rat Irwin test. There were no noticeable
effects on the cardiovascular or respiratory parameters in the anaesthetised dog or any behavioural, autonomic or motor effects in the rat at the doses studied.

Rodent and dog toxicology studies have indicated that the primary target organ of toxicity is the bone marrow with recovery seen following withdrawal of olaparib. *Ex vivo* studies have confirmed that olaparib is cytotoxic to human bone marrow cells.

Olaparib was not mutagenic in the Ames test but was clastogenic in the Chinese hamster ovary (CHO) chromosome aberration test *in vitro*. When dosed orally, olaparib also induced micronuclei in the bone marrow of rats. This profile is consistent with the potential for genotoxicity in man.

Reproductive toxicology data indicate that olaparib can have adverse effects on embryofoetal survival and development at dose levels that do not induce significant maternal toxicity.

Further information can be found in the current version of the olaparib IB.

## 1.1.9 Clinical experience

Clinical experience with olaparib is fully described in the current version of the olaparib IB.

# 1.1.9.1 Olaparib monotherapy studies in breast cancer patients Study D0819C00003

Olaparib demonstrated a statistically significant improvement in PFS in Study D0819C00003 (OlympiAD), a randomised Phase III study comparing olaparib to chemotherapy of physician's choice (TPC) in the treatment of *gBRCAm* HER2 negative metastatic breast cancer. At 77% maturity, PFS by blinded independent central review was significantly longer in patients treated with olaparib vs. TPC (HR 0.58; 95% CI 0.43-0.80; p=0.0009; 7.0 vs 4.2 months, respectively). Results in the East Asian and White sub-populations were consistent with these findings. PFS2 (time to second progression; investigator-assessed) was also longer in the olaparib arm (HR 0.57; 95% CI 0.40-0.83). Objective response rate was 59.9% and 28.8% in the olaparib and TPC arms, respectively. Final analysis of OS at 64% maturity revealed a median OS of 19.3 months for olaparib vs 17.1 months for TPC (HR 0.90; 95% CI 0.66-1.23) (Robson et al 2017).

# Study D0810C00002

Study D0810C00002 was a Phase I open-label, dose escalation and cohort expansion study in 98 patients with solid tumours. Patients in the dose-escalation cohort received olaparib at doses ranging from 10 mg daily to 600 mg twice daily (b.i.d.); whereas all patients in the dose-expansion cohort received olaparib at 200 mg twice daily after the MTD was identified as 400 mg b.i.d. The main tumours by type were ovarian (54 [55.1%]), breast, (13 [13.3%]); colon (5 [5.1%]), prostate (4 [4.1%]) and skin cancers (4 [4.1%]). Overall 23 patients were *BRCA* mutation carriers; of these, 19 patients had *BRCA* mutated ovarian, breast, or prostate cancer and were evaluable for response. Forty-seven percent (9/19) of the patients had an

objective response as defined by Response Evaluation Criteria in Solid Tumors (RECIST), and 63% (12/19) had stable disease for at least 4 months (Fong et al 2009).

#### Study D0810C00008

Study D0810C00008 was a Phase II proof-of-concept study initiated as an open-label, single-arm, international, multicenter study to assess the efficacy and safety of olaparib given orally b.i.d. in patients with gBRCA1 and gBRCA2 mutations and advanced breast cancer. Patients had a median of 3 previous chemotherapy regimens and approximately half of the patients had TNBC. The primary objective was to assess the efficacy of the capsule formulation at 2 different doses of olaparib in terms of ORR (overall response rate) in patients with advanced breast cancer. Patients received olaparib at a dose of 400 mg b.i.d. or 100 mg b.i.d. continuously in 28-day cycles, for multiple cycles, until no further clinical benefit was apparent or the patient was withdrawn from the study. The cohorts were conducted in sequence, the 400 mg b.i.d. group first (n=27) followed by the 100 mg b.i.d. group (n=27). In the ITT analysis set, the confirmed RECIST ORR overall was 11/27 (41%) at 400 mg b.i.d. and 6/27 (22%) at 100 mg b.i.d. Responses were seen in both gBRCA1 and gBRCA2 carriers. Median time to progression was 5.3 months for the 400 mg b.i.d. group and 3.7 months for the 100 mg b.i.d. group (Tutt et al 2010).

#### Study D0810C00020

Study D0810C00020 was a Phase II open-label, non-randomised study of olaparib in patients with known *gBRCA* or high-grade serous/undifferentiated ovarian cancer and patients with known *gBRCA* or TNBC. All patients received olaparib 400 mg b.i.d. until disease progression or until the investigator believed it was in the best interest of the patient to stop treatment. Tumour response data was analysed in 64 ovarian (*BRCA* or serous ovarian) and 26 breast (*BRCA* or triple negative) cancer patients who received olaparib 400 mg b.i.d. Germline *BRCA* mutations were present in 11 of the 26 breast cancer patients. Median number of prior chemotherapies in the breast cancer group was 3 (range: 1 to 7). Over 70% of the breast cancer patients had received 3 or more previous lines of prior chemotherapy, with a median of 35.3 months from diagnosis to start of treatment with olaparib. None of the breast cancer patients achieved a RECIST response. However, 63% of the patients with *BRCA* mutations had an overall best response of SD lasting 8 weeks or more. The median PFS in this cohort was 3.6 months in this group (Gelmon et al 2011).

#### Study D0810C00042

Study D0810C00042 was a Phase II, open label, non-randomised, non-comparative, multicenter study in patients with advanced cancers who had confirmed germline *BRCA1* and/or *BRCA2* mutations. A total of 62 breast cancer patients were recruited, all of whom received at least 3 prior lines of therapy (with a median of 6 prior regimens). Eight (12.9%) of the breast cancer patients had an OR and the median duration of response was 204 days. At 16 = weeks, disease control was observed in 23 (37.1%) patients. The median PFS (progression free survival) was 3.68 months. The median OS was 11.01 months; the survival rate at 6 months was 74.6%, and at 1 year was 44.7% (Kaufman et al 2014).

The details on the pivotal phase II data in ovarian cancer patients as well as olaparib combination with chemotherapy are presented in the Investigator Brochure.

## 1.2 Research hypothesis

Following completion of definitive local and systemic neoadjuvant or adjuvant chemotherapy treatment, giving olaparib tablets 300 mg b.i.d. (twice daily) in the adjuvant setting for up to 12 months in patients with germline *BRCA* mutations and high risk, Stage II-III HER2 negative primary breast cancer has superior efficacy and acceptable tolerability profile as compared with no further treatment. The efficacy in this study will be assessed by the primary analysis of IDFS defined as the time from randomisation to the date of first treatment failure that is loco-regional, distant recurrence, new invasive cancer or death from any cause. Supportive efficacy analyses include assessment of distant disease free survival and overall survival.

# 1.3 Rationale for conducting this study

The aim of the proposed phase III study is to obtain a reliable evaluation of whether olaparib monotherapy following completion of definitive local and systemic neoadjuvant or adjuvant chemotherapy is sufficiently safe and provides clinically meaningful benefit in the proposed indication.

The primary endpoint of the trial is IDFS, defined as the time from randomisation to date of first treatment failure that is loco-regional or distant recurrence or new cancer or death from any cause. IDFS is further detailed according to the standardised STEEP system definition (Hudis et al 2007) as one of the following:

- Ipsilateral invasive breast tumour recurrence (IIBTR): invasive breast cancer involving the same breast parenchyma as the original primary.
- Regional invasive breast cancer recurrence: invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast.
- Distant recurrence: metastatic breast cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer.
- Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
- Contralateral invasive breast cancer.
- Second primary non-breast invasive malignancies (i.e. excluding new in situ carcinomas at any site). Second primary non-breast invasive malignancies include hematologic malignancies and MDS. Squamous or basal cell skin cancers will not be counted as primary endpoint events.

Considering the tendency of TNBCs to metastasise to viscera more often than other types of breast cancer, and knowing the generally incurable nature of those with metastases, a secondary endpoint of DDFS will be measured to support the primary endpoint of IDFS and help characterise the secondary endpoint of OS.

In addition to TNBC, the study will also allow patients with positive hormone receptor status as long as they are HER2 negative, who have a germline *BRCA* mutation and fulfil additional criteria for high recurrence risk (see Section 4.1 Inclusion crit. 3A, 3B, 4b). While events in these patients might not accumulate at the same rate as in *gBRCA*m TNBC, extrapolations from the metastatic setting (Tutt et al 2010) support the expectations that these patients will also benefit from adjuvant olaparib treatment.

In addition, PARP and *BRCA* function has been linked to estrogen and other hormone receptor transcriptional function (Zhang et al 2013; Schiewer et al 2013), supporting the expectation that additive/synergistic effects could manifest when combining hormonal treatments with olaparib in hormone receptor-positive patients with *gBRCA*m status. Recent preclinical data by Nardone et al (2015) indicate that olaparib may enhance endocrine therapy efficacy and circumvents resistance; as a consequence, addition of olaparib to hormonal treatment might confer additional treatment benefits in patients with high recurrence risk.

Hence, hormone-receptor-positive gBRCAm patients will be allowed to receive hormonal treatments at any time during the study. Based on in vitro P450 inhibition and induction data, olaparib would not be expected to alter the PK of standard hormonal therapies used in the adjuvant setting (tamoxifen, aromatase inhibitors with or without ovarian suppression). Based on a preliminary analysis from an ongoing olaparib/hormonal treatment study sponsored by AstraZeneca (Study D081CC00001) there was no indication for clinically relevant drug-drug interaction between olaparib and the anti-hormonal agents tamoxifen, letrozole or anastrozole.

All patients will be followed for local recurrence, distant recurrence (including subsequent sites of recurrence), new cancers and overall survival for a minimum of 10 years, in order to fully describe the long-term impact of adjuvant olaparib therapy.

#### 1.3.1 Rationale for central *BRCA* mutation test at Myriad Genetics, Inc

The FDA has indicated that the *BRCA1* and *BRCA2* mutation assay will need to be approved as a companion diagnostic in the US.

Myriad Genetics, Inc has been chosen as a partner in developing a companion diagnostic for *BRCA1* and *BRCA2* testing because it has extensive experience in *BRCA1* and 2 mutation detection. Myriad keeps the most comprehensive database on *BRCA1* and 2 gene mutations and their clinical relevance. Furthermore, Myriad has an established laboratory infrastructure, which supports high volume testing with turnaround times that can meet the needs of a clinical trial.

#### 1.4 Benefit/risk and ethical assessment

As of 20 March 2015, approximately 3862 patients with ovarian, breast, gastric, pancreatic, and a variety of other solid tumours are estimated to have received treatment with olaparib in AstraZeneca-sponsored, investigator-sponsored, and collaborative group studies and a Managed Access Programme. Olaparib has been given as either monotherapy (an estimated 2327 patients) or in combination with other chemotherapy/anticancer agents (an estimated 1535 patients). Many of these combination studies are ongoing. An estimated 1835 patients to date have received the capsule formulation of olaparib, 27 patients have received both the capsule and tablet formulation, and 2000 patients have received the tablet formulation. Approximately 878 patients have received comparator or placebo across the olaparib development programme.

An analysis of monotherapy data across 13 AstraZeneca sponsored monotherapy studies in 1006 patients with ovarian cancer and other non-ovarian solid tumours who have been given olaparib capsules estimated that 16.0% (161/1006) of patients had been exposed to olaparib capsules for  $\ge 12$  months, 8,3% (84/1006) for >18 months and 4,1% for >24 months at the time of database closure for the respective studies. Twenty one patients (2.1%) had received  $\ge 48$  months of olaparib exposure. From the available data to date, there is no evidence of any unexpected toxicity following long-term olaparib (capsule) monotherapy exposure.

In a Phase I study in ovarian cancer patients (Study DO810C00024) the 300 mg b.i.d. monotherapy tablet regimen was considered to have an acceptable tolerability profile relative to the 400 mg b.i.d. capsule and has been determined to be the recommended olaparib monotherapy tablet dose for future studies with olaparib using the tablet formulation. Olaparib as monotherapy at doses up to 400 mg b.i.d. (capsule formulation) and 300 mg b.i.d. (tablet formulation) is generally well tolerated, with most common AEs including nausea, fatigue, vomiting, and anaemia. There were mainly mild-to-moderate (CTCAE Grade  $\leq$  2) in severity.

In addition, in a small number of patients MDS/AML or pneumonitis have been observed and identified as important risks.

#### **Important Potential Risks**

## Myelodysplastic syndrome/acute myeloid leukaemia

There have been 21 reports of myelodysplastic syndrome (MDS) and/or acute myeloid leukaemia (AML) in patients treated with olaparib as of 20 March 2015; 14 cases in olaparib monotherapy trials and 7 cases in olaparib combination studies with carboplatin and paclitaxel (n=4) or cediranib (n=1), irinotecan and cisplatin (n=2). A total of 3862 patients are estimated to have received olaparib, giving a cumulative incidence of 0.5% for MDS/AML. Two additional reports of MDS have been received from a blinded study (D0816C00002) in which the treatment of the 2 patients (olaparib or placebo) is unknown, and if these patients are considered to have been on olaparib treatment, the estimated incidence would be 0.6%. MDS was also reported for 2 patients who were known to have received placebo or a comparator in the olaparib trial programme (1 patient received placebo in Study D0810C00019 and 1 patient

received liposomal doxorubicin in Study D0810C00012). The 21 olaparib-treated patients and two patients on blinded treatment had primary ovarian, peritoneal, fallopian tube cancer (n=20), pancreatic cancer (n=2) or breast cancer (n=1) and 18 of them had germline BRCA1/2 mutations (3 cases BRCA status unknown; 2 cases negative). It has been hypothesised that a deficiency in the expression of BRCA genes may leave patients more vulnerable to the adverse effects of chemotherapy, and therefore, at an increased risk of MDS/AML as a result of cancer treatment (Cole and Strair 2010). Eleven patients had received olaparib for  $\leq$  12 months (5 patients had  $\leq$  6 months exposure, 6 patients had 6 to 12 months exposure) and the other 12 cases occurred following longer than 12 months olaparib exposure (2 patients following 12-18 months exposure, 2 patients 18-24 months and 8 patients following  $\geq$  2 years exposure to olaparib).

The median time to onset of t-AML from ovarian cancer diagnosis is reported as approximately 5.5 years (Gupta et al 2007; Vay et al 2011). The overall standardised incidence ratio (8.68 overall) varies over time - 12.07 within 1 to 5 years, 10.81 within 5 to 10 years and 2.30 after 10 years (Morton et al 2013).

Eighteen of the 23 patients died: in 12 of these patients, MDS/AML or myelodysplasia was recorded as either a primary or secondary cause of death. The other 6 deaths were reported as follows: 1 due to cerebral haemorrhage and disseminated intravascular coagulation, 1 due to complication of double umbilical cord blood transplantation and 4 due to disease progression (2 ovarian cancer, 1 breast cancer [patient had a prior history of ovarian cancer treated with platinum-based chemotherapy] and 1 pancreatic cancer). In 5 patients, the event of MDS/AML is reported as ongoing as of the 20<sup>th</sup> March 2015. All patients had other potential features that may be contributing factors for the development of MDS/AML. All patients had received previous chemotherapy with DNA damaging agents including platinum, with many patients having extensive previous chemotherapy with multiple treatment regimens over multiple years including carboplatin, taxanes, anthracyclines, other alkylating and DNA damaging agents and radiotherapy.

Since bone marrow is known to be a target organ for olaparib toxicity, increased risk of MDS/AML with long-term exposure to olaparib cannot be excluded. However, there is insufficient data at present to evaluate this relationship. Moreover, while non-clinical data suggest bone marrow progenitor cell populations are reduced temporarily following olaparib treatment, there is no evidence to date linking olaparib treatment to the generation of abnormal bone marrow precursors. Furthermore, all patients who developed MDS/AML had extensive prior chemotherapy and while it is not possible to exclude the contribution of olaparib, it must be considered that there were other potential contributing factors in all cases. Preclinical data also suggest potential benefit with PARP inhibitors in MDS/AML and clinical trials are now underway to assess this effect (Gaymes et al 2008). The risk of developing MDS/AML as a long term toxicity in breast cancer patients with stage I-III disease exposed to standard dose adjuvant chemotherapy including alkylator and anthracycline with or without taxane, is estimated to be around 0.5% varying between 0.37% and 1.16% (Praga et al 2005, Smith et al 2003, Hershman et al 2007, Burnell et al 2010, Aebi et al 2011). Both alkylators and

topoisomerase II inhibitors (anthracyclines) have been associated with treatment related MDS/AML. The risk is perceived as low and not outweighing the benefit of adjuvant chemotherapy in breast cancer patients. To ensure robust safety monitoring, patients in this clinical trial will have safety assessments every two weeks during the first month and monthly safety assessments for the first 6 months of treatment followed by 3 monthly assessments until completion of treatment (maximum 12 months treatment). In addition, an Independent Data Monitoring Committee (IDMC) will review the emerging safety data from the trial in an unblinded fashion. Long term safety follow-up will be implemented in the trial. Clinical guidelines for managing bone marrow toxicity are implemented as part of the safety management plan (Section 5.5.6).

#### **Pneumonitis**

As of 20 March 2015, 14 patients out of a total of 3862 patients, estimated to have received olaparib, have reported pneumonitis, giving a cumulative incidence of 0.36% for pneumonitis. Six additional reports of pneumonitis have been received from 4 blinded studies, where the treatment of the patients is unknown (3 either olaparib or placebo; 2 either olaparib + paclitaxel or placebo + paclitaxel and 1 olaparib + abiraterone or placebo + abiraterone). If these patients were considered to have been on olaparib treatment, the estimated cumulative incidence would be 20/3862 (0.52%). Pneumonitis was also reported for 2 patients (1%) of 190 patients that received placebo or comparator in the olaparib trial programme (1 patient on placebo in Study 19 and 1 patient on paclitaxel in Study 39). The patients were treated with olaparib for breast cancer (n=3), ovarian cancer (n=6), non-small cell lung cancer (NSCLC) (n=4), small cell lung cancer (SCLC) (n=1), pancreatic cancer (n=1), gastric cancer (n=3), prostate cancer (n=1) and thymic cancer (n=1). The reports of pneumonitis presented with no consistent clinical pattern and were heavily confounded by a number of pre-disposing factors (including disease under investigation, underlying pulmonary disease, pre-existing medical conditions, smoking history and/or previous chemotherapy and radiotherapy). The majority of patients had received prior radiotherapy and/or chemotherapy and had other risk factors within the medical histories including pneumonitis, interstitial lung fibrosis, dyspnoea, haemoptysis, chest infection, allergic asthma, pleural effusion, pleural metastases and smoking. Five patients had current SCLC or NSCLC. An independent review of available chest computed tomography (CT) scans and radiographs associated with the reports of pneumonitis concluded that there appeared to be no clear consistent clinical pattern.

Investigation of any new or worsening pulmonary symptoms has been implemented as part of the safety management plan (Section 5.5.6).

## New Primary Malignancies other than MDS/AML

Overall, the number of reports of new primary malignancies is low, with 24 events (in 22 patients) being reported to 20 March 2015 in 3862 olaparib treated patients (0.57%) and one event (bladder cancer) reported in the placebo arm of the double-blind Study 19. Three additional reports of new primary malignancies have been received from 1 blinded study for the maintenance treatment of ovarian cancer (D0818C00001, tablet formulation), where the

treatment of the patients is unknown (either olaparib or placebo). If these patients are considered to have been on olaparib treatment, the estimated cumulative incidence would be 0.65%.

The types of new primary malignancies reported in the 22 patients on olaparib treatment were breast cancer, colon cancer, lung neoplasm malignant, gastric cancer, plasma cell myeloma, basal cell carcinoma, skin cancers, neoplasm skin, squamous cell carcinoma, malignant melanoma, malignant muscle neoplasm, precursor T-lymphocytoc lymphoma/leukaemia, tongue cancer and papillary thyroid carcinoma. The 3 patients on blinded treatment reported new primary breast cancer malignancies.

Of the 25 patients (22 on olaparib, 3 on blinded treatment) subsequently diagnosed with a new primary malignancy, the majority were reported whilst receiving study treatment (21 patients). In 4 patients the event was reported after olaparib discontinuation (within 60 days after olaparib discontinuation in 2 patients, and more than 240 days after olaparib discontinuation in 2 patients).

The duration of treatment for the 25 patients was:

- <6 months for 5 patients
- 6 to 12 months for 8 patients
- 12 to 18 months for 2 patients
- 18 to 24 months for 3 patients
- >2 years for 7 patients.

The type of new primary cancers reported were generally in line with secondary cancers observed in ovarian and breast cancer populations reported in the literature (Bergfeldt et al 1995, Fowble et al 2001, Wesolowski et al 2007), or were cancers such as skin cancer, known to be the most common cancer in the general population and associated with high cure rates.

Ovarian cancer patients have been reported to have an increased risk of developing second primary malignancies. Patients with germline *BRCA* mutations are at risk of developing other primary cancers notably breast cancer. Ginsburg et al 2010 reported higher rates of skin cancers in patients with *BRCA1* (1.6%) and *BRCA2* (3.0%) mutations.

There were other contributing factors/potential alternative explanations for the development of the new primary malignancy in all 22 olaparib treated patients and the 3 on blinded treatment. All patients had previously received various chemotherapy agents including multiple cycles of DNA damaging platinum containing chemotherapies, taxanes, anthracyclines and other alkylating and DNA damaging agents. Four patients were reported to have had prior radiotherapy. Twenty two patients had a documented breast cancer gene mutation (*BRCA* 1

or 2). Seven of the 25 patients had previous medical histories of cancer (ovarian, cervix, breast, peritoneal) and 3 patients with skin cancers either had previous basal cell carcinoma reported or skin lesions evident prior to study treatment.

There is insufficient evidence for an association between olaparib treatment and the development of new primary malignancies in the clinical trial programme to date. The risk is perceived as low and not outweighing the benefit of adjuvant chemotherapy in breast cancer patients. An IDMC will review the emerging data from the trial in an unblinded fashion.

#### Potential benefit

A Marketing Authorisation Application was approved in EU/EEA on 16 December 2014 for the indication 'LYNPARZA monotherapy for the maintenance treatment of adult patients with platinum-sensitive relapsed BRCA-mutated (germline and/or somatic) high grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in response (complete response or partial response) to platinum-based chemotherapy.'

A New Drug Application was approved in the US on 19 December 2014 for the indication 'LYNPARZA monotherapy in patients with deleterious or suspected deleterious germline BRCA mutated (as detected by an FDA-approved test) advanced ovarian cancer who have been treated with three or more prior lines of chemotherapy.'

Olaparib tablet formulation was approved in January 2018 for patients with deleterious or suspected deleterious *gBRCAm*, HER2-negative metastatic breast cancer who have previously been treated with chemotherapy in the neoadjuvant, adjuvant or metastatic setting. Patients with hormone receptor-positive breast cancer should have been treated with a prior endocrine therapy or be considered inappropriate for endocrine treatment.

Phase II clinical studies have investigated the effect of olaparib either as monotherapy or in combination with other chemotherapy agents in cancer patients. In patients carrying germline BRCA mutations, monotherapy studies in patients with heavily pre-treated breast cancer have reported an ORR of up to 41%.

In ovarian cancer patients, the pivotal phase II study D0810C00019, a double-blind, randomised study assessed the efficacy of olaparib 400 mg b.i.d capsules as a maintenance treatment following platinum-based chemotherapy in patients with platinum sensitive relapsed high grade serous ovarian cancer. The PFS following olaparib maintenance therapy was significantly longer compared with the placebo group (HR 0.35; 95% CI: 0.25, 0.49; p<0.00001) in the overall population. In the subgroup of patients with *BRCA* mutant ovarian cancer, the effect was even greater with a PFS HR of 0.18 (95% CI: 0.11, 0.31; p<0.00001; median 11.2 versus 4.3 months). An interim analysis of OS was performed at 58% maturity. In the overall population, the analysis demonstrated a non-statistically significant numerical advantage for olaparib-treated patients (OS HR 0.88; 95% CI 0.64-1.21; p=0.43808) and there was again a greater effect in the *BRCA*-mutated subgroup: the OS HR was 0.74 (95% CI 0.46 to 1.19; p=0.20813) with a numerical advantage in median OS observed with olaparib (median

34.9 months versus 31.9 months with placebo). Among the 62 placebo-treated patients with *BRCA* mutations, 14 switched to a PARP inhibitor post progression.

Based on these results and data from the full clinical program to date, it is anticipated that in the adjuvant setting, olaparib will have a positive benefit risk profile for the treatment of the small well-defined population of high-risk HER2 negative primary breast cancer patients with *BRCA* mutations.

#### 2. STUDY OBJECTIVES

# 2.1 Primary objective

The primary objective is to assess the effect of adjuvant treatment with olaparib on Invasive Disease Free Survival (IDFS).

# 2.2 Secondary objectives

The secondary objectives of this study are:

- 1. To assess the effect of adjuvant treatment with olaparib on overall survival (OS)
- 2. To assess the effect of adjuvant treatment with olaparib on Distant Disease Free Survival (DDFS)
- 3. To assess the effect of adjuvant treatment with olaparib on the incidence of new primary contralateral breast cancers (invasive and non-invasive), new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer
- 4. To assess the effect of olaparib on patient reported outcomes using the FACIT-Fatigue and EORTC QLQ-C30 questionnaires
- 5. To assess the efficacy of olaparib in patients identified as having a deleterious or suspected deleterious variant in either of the *BRCA* genes using variants identified with current and future *BRCA* mutation assays (gene sequencing and large rearrangement analysis)
- 6. To determine the exposure to olaparib (in plasma) in patients receiving olaparib as adjuvant therapy

# 2.3 Safety objective

To assess the safety and tolerability of adjuvant treatment with olaparib





# 3. STUDY PLAN AND PROCEDURES

This Clinical Study Protocol has been subject to peer review according to AstraZeneca standard procedures.

# 3.1 Overall study design, flow chart and study schedules

This is a randomised, double-blind placebo controlled multicentre, phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy.

Randomised patients will receive study treatment for up to a maximum of 12 months. All patients will have safety assessments every 2 weeks during the first month, every 4 weeks for the following 5 months (up to week 24) and 3 monthly for the remaining 6 months of study treatment, plus 30 days after its discontinuation. Efficacy assessments (medical history and physical examination) will be performed on a 3 monthly basis during the first 2 years following end of study treatment, followed by 6 monthly assessments for years 3, 4 and 5 and annually thereafter. Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory before enrolment (within 12 months prior to Screening PART 1) and during study participation (starting at week 24 and yearly thereafter) for patients with any remaining intact breast tissue (including male patients). The preferred tests are mammogram or magnetic resonance imaging (MRI; MRI preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion. Evidence of disease recurrence or new primary cancer will require histopathological and/or radiological confirmation

Patients who develop loco-regional recurrence should have cytological/histological confirmation. Loco-regional recurrence should be treated with curative intent when possible. Appropriate imaging (CT, MRI bone and/or PET scan) of the chest/abdomen/pelvis or any other area as clinically indicated (MRI preferred to examine CNS (central nervous system) if new neurological symptoms occur) should be performed at the time of local recurrence to exclude further spread of the disease.

Distant recurrence should be diagnosed by radiological/imaging examination and every attempt should be made for histopathological confirmation when metastatic lesion is accessible for biopsy.

If the patient meets the IDFS endpoint due to a breast cancer related distant relapse, the patient will enter the survival follow-up phase of the trial, with annual assessments from the date of distant relapse, which will continue until 10 years after the last patient is randomised. No clinic visits will be required during the survival follow-up phase; information may be collected via telephone, medical records or death registries. During the survival follow-up phase, in addition to vital status, the following information will be collected (if available): specific cancer therapies (only first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time), sites of metastases and any other new cancers.

If the IDFS endpoint is met due to events other than distant relapse, the patient will continue the efficacy assessment visit study schedule until breast cancer related distant relapse occurs, or approximately 10 years following their randomisation into the study, whichever occurs first. They will then enter the survival follow-up phase of the trial.

See Section 5.8.1 for guidelines on study visits for any patient discontinuing prior to completing 52 weeks of study treatment.

#### Figure 1 Study Flow Chart

ICF for patients with unknown BRCA status to undergo central BRCA testing during, or prior to, neoadjuvant/adjuvant chemotherapy



by 6 monthly assessments for the 3rd, 4th and 5th year, and annually thereafter

Yearly breast imaging (mammogram and/or MRI) (ipsilateral and/or contralateral) for 10 years\*

\*The study will end 10 years after the last patient has been randomised

#### Figure 2 Screening Plan

# Screening PART 1– Patients with Unknown gBRCA Mutation Status:

• Only those patients who **do not** know their gBRCA mutation status prior to entry in to the study

These patients will undergo screening assessments as described for PART 1 in Table 1. Screening PART 1 is conducted to determine if the patient is considered **eligible to undergo the** *BRCA* **status blood test**. Once PART 1 has been successfully completed and patients have had a *BRCA* test, these patients will continue to PART 2 and have all procedures performed as described for PART 2 (see Table 1)

## Screening – PART 2 – ALL Patients (Patients with Known gBRCA Mutation Status):

- Those patients who already know their gBRCA mutation status **and** have a deleterious or suspected deleterious mutation to undergo screening assessments as described for PART 2 (see Table 1)
- Those patients originally with unknown gBRCA status who have completed screening PART 1 and now have a confirmed deleterious or suspected deleterious mutation should undergo screening assessments as described for PART 2 (see Table 1)

Table 1 Study Schedule - Screening (PART 1 and PART 2)

| Day | Any time prior, during or after neoadjuvant/adjuvant chemotherapy or radiotherapy PART 1 a (ONLY Patients requiring a gBRCA status Myriad test before randomisation) | -28 to 0 days PART 2 (Patients with confirmed gBRCA status by Myriad or if BRCA status is known prior to study entry <sup>j</sup> ) |
|---|---|---|
| Informed consent | X bc | X <sup>j</sup> |
| Demographics (date of birth) | X | X |
| Medical and surgical history d | | X |
| Prior cancer therapies including radiotherapy | | X |
| Inclusion/exclusion criteria | X (all ** criteria) | X |
| ECOG Performance Status | | X |
| Physical examination | | X |
| Vital signs | | X |
| ECG <sup>f</sup> | | X <sup>g</sup> |
| Haematology / clinical chemistry/Coagulation ° | | X |
| Urinalysis <sup>h</sup> | | X |
| Pregnancy test i | | X |
| EORTC QLQ-C30 n | | X |
| FACIT-Fatigue <sup>n</sup> | | X |
| Blood sample for determination of <i>BRCA</i> status via Myriad | X | X e |
| Blood sample for assessment of current and future <i>BRCA</i> mutation assay(s) <sup>c</sup> | X | X e |
| Concomitant medications | | X |
| Archival tumour sample (FFPE) (mandatory) k | | X |
| Surgical tumour sample (FFPE) (post neoadjuvant chemotherapy (mandatory)) k | | X |

# Table 1 Study Schedule - Screening (PART 1 and PART 2)

| Day | Any time prior, during or after neoadjuvant/adjuvant chemotherapy or radiotherapy PART 1 a (ONLY Patients requiring a gBRCA status Myriad test before randomisation) | -28 to 0 days PART 2 (Patients with confirmed gBRCA status by Myriad or if BRCA status is known prior to study entry <sup>j</sup> ) |
|---|---|---|
| Radiological assessment to exclude metastatic breast cancer (where applicable) <sup>1</sup> | | X |
| Family history of cancer | | X |
| Serious Adverse Events <sup>m</sup> | X (only SAEs due to study procedures) | X (SAEs only) |

- a The time period is to allow those patients that require a Myriad gBRCA sample to have the test taken and the results returned prior to randomisation.
- b It is recommended that patients that require the Myriad gBRCA sample testing are to be consented for BRCA testing and participation in the trial prior or during neoadjuvant/adjuvant chemotherapy prior to entering the study.
- c Any patient who consents to study related Myriad gBRCA status testing, must also have a blood sample taken at the same time for the purpose of developing and validating a future mutation assay.
- d Include history of blood transfusion within previous 120 days from start of study treatment and the reasons e.g. bleeding. Additionally CPS+EG score components should be collected (Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS)) for the non-pCR patients who received prior neoadjuvant chemotherapy. Instructions on how to calculate the CPS&EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix H.
- e Samples to be taken in screening PART 2 only for patients with known gBRCA mutation who have not completed PART 1.
- f ECG recordings should be performed once the patient has been in the supine position for at least 5 minutes
- ECG assessments to be completed within 28 days before randomisation.
- h Urinalysis (dipstick) should be performed at screening. After screening, urinalysis will only be required if clinically indicated.
- i Women who are not postmenopausal or have not undergone hysterectomy must have a negative urine or serum pregnancy test within 28 days prior to randomisation and a confirmatory test on Day 1 before starting study treatment. If results are positive the patient is ineligible.
- j Patients for whom their gBRCA status is already known, should be consented to the study within 28 days prior to randomisation.
- Mandatory for all randomised patients i.e. for adjuvant patients this refers to the surgical specimen; for neoadjuvant patients, both the pre-treatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required. Samples will only be sent to the study bio-repository once the patient has been randomised.

Patients considered at high risk of having disseminated disease (i.e. those with locally advanced disease, clinical N2-3 or pathological N1-3 with the exception of pN1a in adjuvant patients are expected to have a CT/MRI scan of the Thorax/Abdomen/Pelvis or any other area as clinically indicated and a bone scan at any point between diagnosis of the current breast cancer and randomisation to rule out metastatic breast cancer. (Note PET/CT scan may be used as an alternative imaging technique and precludes the need for bone scan). Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory before enrolment (within 12 months prior to Screening PART 1) for patients with any remaining intact breast tissue (including male patients). The preferred tests are mammogram or MRI (MRI preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion.

To rule out metastatic breast cancer, patients with screening ALT/AST or ALP above institutional upper limit of normal should have liver ultrasound, CT or MRI at any time point between diagnosis of current breast cancer and randomisation. Screening bone scan is required if ALP and/or corrected calcium level are above the institutional upper limit. (Note PET/CT scan may be used as an alternative imaging technique).

- m Serious adverse events must be captured from time of consent. In Screening PART 1 of the study only SAEs related to a study procedure will be collected. In Screening PART 2 all SAEs will be collected.
- n EORTC QLQ-C30 + FACIT-Fatigue will be collected prior to randomisation once eligibility is confirmed.
- o Coagulation analysis only required at baseline.

Study Schedule - On treatment (Year 1)

Table 2

| Visit Number | 2 | ю | 4 | 5-9<br>(Every 4<br>weeks) | 10-11<br>(Every 3<br>months (14<br>weeks)) | Premature study<br>treatment<br>discontinuation <sup>g</sup> | Follow-up 30 days after last dose of study medication (all patients) |
|---|---|---|---|---|---|---|---|
| Week | 0 | 2 | 4 | 8, 12, 16, 20, 24 | 38, 52 | | |
| Day | 1 | 15 | 29 | | | | |
| Visit Window | | р€∓ | р€∓ | ±1 week | ±2 week | +2 week | +2 week |
| Serum or urine pregnancy test for women of childbearing potential <sup>a</sup> | X | | X | X | X | | X |
| ECOG performance status | q X | | | | | | |
| Vital signs | q X | | X | X (weeks 12 and 24 only) | X | X | X |
| Haematology / clinical<br>chemistry ° | Х р, с | X | X | X | X | X | X |
| Recurrent/new cancers assessment (includes physical exam <sup>d</sup> , clinical signs and symptoms) | X | | | X (weeks 12 and 24 only) | Х | Х | X |
| Mammogram and/or breast<br>MRI (ipsilateral and/or<br>contralateral) (MRI<br>preferred for patients<br>younger than 50 years) <sup>e</sup> | | | | X (week 24 only) | | | |
| Adverse Events | X | X | × | X | X | X | X |

Study Schedule – On treatment (Year 1)

Table 2

| Visit Number | 7 | e | 4 | 5-9<br>(Every 4<br>weeks) | 10-11<br>(Every 3<br>months (14<br>weeks)) | Premature study treatment discontinuation § | Follow-up 30 days after last dose of study medication (all patients) |
|---|---|---|---|---|---|---|---|
| Week | 0 | 2 | 4 | 8, 12, 16, 20, 24 | 38, 52 | | |
| Day | 1 | 15 | 29 | | | | |
| Visit Window | | ±3d | ±3d | ±1 week | ±2 week | +2 week | +2 week |
| Concomitant medications including blood transfusions | × | × | × | × | × | X | X |
| Demographics <sup>j</sup> | × | | | | | | |
| EORTC QLQ-C30 | | | | X (week 24 only) | X (week 52 only) | | |
| FACIT-Fatigue | | | | X (week 24 only) | X (week 52 only) | | |
| Biomarker Blood 2 samples (mandatory) | × | | | | | | X |
| PGx Blood sample (optional) | X | | | | | | |
| Blood sample for PK<br>analysis (optional; after<br>signing PK Informed<br>consent) (subset of<br>patients) <sup>h</sup> | | | × | | | | |

Study Schedule – On treatment (Year 1)

Table 2

| Visit Number | 7 | 3 | 4 | 5-9<br>(Every 4<br>weeks) | 10-11<br>(Every 3<br>months (14<br>weeks)) | reatment days after last discontinuation green medication (a medication (a patients) | Follow-up 30<br>days after last<br>dose of study<br>medication (all<br>patients) |
|---|---|---|---|---|---|---|---|
| Week | 0 | 2 | 4 | 8, 12, 16, 20, 24 38, 52 | 38, 52 | | |
| Day | 1 | 15 | 29 | | | | |
| Visit Window | | р€∓ | р€∓ | ±1 week | ±2 week | +2 week | +2 week |
| Blood biomarker samples<br>at disease recurrence<br>(Mandatory) | × | X | X | × | × | X | X |
| Tumour sample at disease recurrence (Optional) <sup>k</sup> | × | X | × | × | X | X | X |
| Olaparib<br>dispensed/returned <sup>f</sup> | X | | X | X | X | X | |

Pregnancy tests on serum or urine samples will be performed for women of childbearing potential within 28 days prior to randomisation, on Day 1 of the study prior to commencing treatment, at the time points shown in Table 2 during study treatment and at the 30 day follow up visit. If results are positive the patient is ineligible/must be discontinued from study treatment immediately. Details of the pregnancy tests must be recorded in the patient's medical If assessed within 7 days before randomisation, it does not need to be repeated on Day 1 of study treatment unless investigator believes that it is likely to have changed significantly.

Safety blood samples do not need to be repeated on Day 1 of study treatment if they have been assessed within 7 days before randomisation and which significantly. Safety blood samples are to be collected every 2 weeks during the first 4 weeks, then every 4 weeks until week 24 and then at weeks 38 must have been done at least 3 weeks after the last dose of chemotherapy, unless the investigator believes that they are likely to have changed and 52 of study treatment.

reatment is discontinued (data is not required to be captured on an eCRF, however any significant changes from baseline must be reported as an AE). Physical examination both local and general should be performed at day 1 and then at weeks 12, 24 and 38 and 52 post randomisation until study

24 and yearly thereafter) for patients with any remaining intact breast tissue (including male patients). The preferred tests are mammogram or MRI (MRI Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory during study participation (starting at week preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical

examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion.

Sufficient study treatment should be dispensed for at least each treatment period plus overage, however additional treatment can be dispensed to patients to last longer in accordance with local practice.

ad

- regimens containing PARP inhibitors or platinum received by the patient at any time), sites of metastases and any other new cancers. If a recurrent/new followed by the 30 day follow-up visit and site staff completes relevant CRF pages as required. In case of premature treatment discontinuation only the first. They will then enter the survival follow-up phase of the trial. During the annual survival follow-up phase, in addition to vital status, the following distant relapse and until 10 years after the last patient is randomised. If the IDFS endpoint is met due to other events, the patient will continue the study visits where efficacy assessments are scheduled should be performed i.e. week 12, 24, 38, 52 (as applicable) in Year 1 and all visits in Year 2 onwards. cancer assessment is scheduled within 4 weeks of the study treatment discontinuation visit it can be performed at the 30-day follow-up visit (for more schedule until a breast cancer related distant relapse occurs or approximately 10 years following their randomisation into the study, whichever occurs therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse. The date of If a patient discontinues prior to completing 52 weeks of study treatment, the patient should have the study treatment discontinuation visit performed Collection of vital signs, AEs, haematology/clinical chemistry results and concomitant medications is no longer required. Information on endocrine endpoint is met due to breast cancer related distant relapse, the patient enters the survival follow-up phase and is assessed annually from the date of subsequent regimens containing PARP inhibitors or platinum received by the patient at any time) should also be recorded on the eCRF. If the IDFS nformation will be collected (if available): specific cancer therapies (only first line treatment for first breast cancer recurrence and any subsequent discontinuation, the reasons, and details of the following specific cancer therapies (first line treatment for first breast cancer recurrence and any details see Section 5.8.1).
- following sampling windows: 0 to 0.5 h post dose, >0.5 to 1.5 h post dose, 3 to 6 h post dose and >6 to 12 h post dose (before evening dose) preferably on visit 4, day 29. Nevertheless, the samples can also be taken at a later treatment visit, provided that PK consent was obtained beforehand (for details PK sampling (optional) to be performed in a subset of patients. Sampling times: pre-dose (before morning dose) plus one sample in each of the P
- Blood samples (plasma and serum) for biomarker analysis should be collected on Day 1 prior to first dose of study treatment.
  - j Race and ethnicity data to be collected unless not allowed by local regulations.
- The provision of tumour tissue is encouraged only if clinically appropriate and not considered detrimental to patient care and patient signed the appropriate consent form.

Study Schedule - Follow-up Visits (Year 2 onwards)

Table 3

| Month 15 18 21 24 30 36 42 48 Visit Window ±1month ±1month ±2months Recurrent/new cancers assessment (includes physical exam, clinical signs and symptoms) X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | 12 13 14 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | Survival<br>Follow-up<br>(Every 12<br>months) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 15 18 21 24 30 36 | 2 | 3 | | 4 | | S | | 9 | 7 | <b>∞</b> | 6 | 10 | 11+ |
| sical X X X X X X X X X X X X X X X X X X X | 18 21 | 30 | | | 48 | 54 | 09 | 99 | 78 | 06 | 102 | 114 | 126, 138,<br>etc. |
| sical X X X X X X X X X X X X X X X X X X X | ±1month | | + | -2mor | ıths | | | | +1 | ±3months | ths | | ±3months |
| rred | X | × | | | | × | × | × | X | X | X | X | |
| assessment | X | × | | × | | × | | × | × | × | × | × | |
| assessment | X | × | | | | × | × | × | × | × | X | X | $X^{q}$ |
| 30 | | | | | | | | | | | | | $X^{\mathrm{d}}$ |
| r samples at X X X X X X X X X X X X X | | | | | | | | | | | | | |
| amples at X X X X X X X | | | | | | | | | | | | | |
| (Mandatory) | X | | | | | × | × | × | × | × | X | X | |

| Visit Number | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | 12 13 14 15 16 17 18 19 20 21 22 23 24 25 26 Survival Follow-up (Every 12 months) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Year | | 7 | | | 3 | • | 4 | | S | | 9 | 7 | 8 | 6 | 5 6 7 8 9 10 | 11+ |
| Month | 15 | 18 | 21 | 24 | 30 | 36 | 42 | 48 | 54 | 09 | 99 | 78 | 06 | 102 | 114 | 15 18 21 24 30 36 42 48 54 60 66 78 90 102 114 126,138, etc. |
| Visit Window | | ±1month | onth | | | | ±2months | nths | | | | # | ±3months | ths | | ±3months |
| Tumour sample at disease recurrence (Optional) ° | X | X | X | X | X | X | X | X | X | X | X | X | × | X | X | |
| $\mathrm{SAE}^{\mathrm{e}}$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X | x x x x x x x x x x x x x x x x x x x | X |

24 and yearly thereafter) for patients with any remaining intact breast tissue (including male patients). The preferred tests are mammogram or MRI (MRI Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory during study participation (starting at week examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical clinical exam may be supplemented by ultrasound exams at investigator's discretion.

time need to be recorded. Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to First line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any breast cancer related distant relapse.

During the survival follow-up phase, information (where available) on further subsequent cancer therapies (see footnote b), sites of metastases and any The provision of tumour tissue is encouraged only if clinically appropriate and not considered detrimental to patient care and patient signed the appropriate consent form.

followed to resolution unless the event is considered by the investigator to be unlikely to resolve, or the patient is lost to follow-up or in survival followperiod should be reported as an SAE. Non-melanoma skin cancers need to be reported as a non-serious AE unless at least one of the seriousness criteria AstraZeneca Patient Safety according to SAE reporting procedures for this study, regardless of investigator's assessment of causality or knowledge of he/she considers there is a reasonable possibility that the event is causally related to the study treatment, the investigator should report it according to up. If an Investigator learns of any SAEs, including death, at any time after a patient has completed the 30 days post treatment follow-up period, and All ongoing AEs/SAEs and any new AEs/SAEs identified during the 30 calendar days follow-up period after last dose of study medication must be SAE reporting procedures for this study. Any cases of MDS/AML, new primary malignancies or pneumonitis occurring after the 30 day follow-up he treatment arm. If a patient develops MDS/AML full diagnostic details and classification should be provided e.g. bone marrow and cytogenetic s met which then requires to be reported as an SAE, see Section 6.4.2. Any of these types of serious or non-serious events need to be reported to other new cancers will be collected in addition to vital status.

analysis reports, see Sections 5.5.6.3 and 6.4.5.5. A questionnaire will be sent to any investigators reporting MDS/AML or new primary malignancies as an aid to provide detailed information on the case.

# 3.2 Rationale for study design, doses and control groups

#### 3.2.1 Rationale for study design

In this placebo-controlled, double-blinded adjuvant study, TNBC patients and ER and/or PgR positive HER2 negative patients with germline *BRCA* mutations at high risk of recurrence will be randomised to receive monotherapy olaparib 300 mg tablet b.i.d. (twice daily) or corresponding placebo for a maximum of 12 months following completion of their definitive loco-regional treatment and chemotherapy in the adjuvant or neoadjuvant setting.

The rationale for allowing patients with ER and/or PgR positive HER2 negative breast cancer who carry a *gBRCA*m (including gene rearrangements) is provided in Section 1.3.

The use of a placebo comparator to olaparib is considered acceptable in order to objectively test the hypothesis of improved efficacy with the addition of olaparib for up to 12 months as compared to no further therapy (i.e. placebo) in patients with TNBC and endocrine therapy alone in patients with ER and/or PgR positive cancer. By blinding patients and investigators, using placebo control and assessing patients for disease recurrence at pre-defined intervals, the risk of bias that could affect the interpretation of the IDFS endpoint should be minimised. In line with international clinical guidelines evidence of disease recurrence will be assessed during the regular follow-ups (3 monthly during the first 2 years, 6 monthly during the 3rd, 4th and 5th year and annually afterwards) by medical history, physical examination and mammogram and/or breast MRI (MRI preferred for patients younger than 50 years) (ipsilateral and/or contralateral), unless clinical signs and symptoms require further investigation (Khatcheressian et al 2012). In addition safety follow-ups are implemented during the 12-month study treatment period and 30 days after its discontinuation.

It should be noted that the safety and efficacy of olaparib has been demonstrated in the clinical program using the capsule formulation (400 mg - 8 capsules - twice daily); however, an improved tablet formulation (2 tablets twice daily) has been developed and will be used in this study. The tablet dose of olaparib that will be investigated is 300 mg b.i.d. (twice daily) which is considered similar to the capsule 400 mg b.i.d. (twice daily) dose. This tablet dose has been chosen based on data from Study D0810C00024. Since it has been shown that the capsule and tablet formulations are not bioequivalent, a formulation switch based on bioequivalence has not been possible. The tablet dose of 300 mg b.i.d. is considered to have similar efficacy in terms of tumour shrinkage in ovarian cancer patients with *BRCA* mutations to the 400 mg b.i.d. capsule. The 300 mg b.i.d. tablet dose matches or exceeds the exposure of the 400 mg capsule in terms of AUC, C<sub>maxss</sub>, and C<sub>minss</sub>. The tolerability profile of the 300 mg b.i.d. tablet dose in Study D0810C00024 was considered similar to the 400 mg b.i.d. capsule formulation. The most common AEs were consistent with the known safety profile of olaparib, namely low grade nausea, vomiting, fatigue, and anaemia. Further information is provided in the olaparib Investigator's Brochure.

## 3.2.2 Rationale for patient reported outcomes

The patient population for this study will have had intensive treatments with chemotherapy (neoadjuvant or adjuvant), surgery, and possibly radiation therapy prior to entry and randomisation on this study. Prior research by the NSABP and other investigators has demonstrated physical disruption and many symptoms at the end of primary treatment (Ganz et al 2011B, Ganz et al 2004). Research has shown that it may take a year or more for the physical and emotional recovery and that symptoms may persist well beyond improvements in health related quality of life (HRQoL) (Ganz et al 2011A, Ganz et al 1998A, Ganz et al 1998B, Ganz et al 2002, Bower et al 2000, Bower et al 2006). Thus, in any studies that are designed to capture patient-reported outcomes (PROs) of treatment, consideration should be given to assessment of both HRQoL and symptoms.

In this trial of olaparib versus placebo, there is an important opportunity to determine whether or not the use of olaparib delays or retards recovery after primary breast cancer treatment, and if so, what aspects of symptoms and HRQoL are impaired. Gelmon et al 2011 reported on a Phase II open label study of olaparib in breast and ovarian cancer patients, in which fatigue was the most common reported toxicity (50-70% of patients) followed by nausea (62-66%), vomiting (35-39%), and decreased appetite (27-36%). In a Phase II study in patients with *BRCA1* or *BRCA2* mutations and advanced breast cancer, fatigue was the most significant toxicity (41% grade 1-2, and 15% grade 3-4) in the cohort given olaparib 400 mg twice daily (Tutt et al 2010). These trials did not use PROs, and since they were conducted in patients with advanced disease, there is uncertainty about how much fatigue patients will have in the B-55/6-13 trial. However, since this is the most frequent side effect of olaparib, it is our primary patient reported outcome in this placebo-controlled comparison.

The FACIT-Fatigue scale will be used to measure treatment related fatigue. The FACIT-Fatigue measure that is being used in this study is well-established and available in multiple languages.

A standard measure of health-related cancer specific HRQoL, the EORTC QLQ-C30, will be used in this study to track recovery in key domains of HRQoL in the year after initial treatment, and to measure symptoms, with a heightened focus on fatigue and GI symptoms (nausea, vomiting, diarrhea), as these symptoms have been reported with olaparib. The GI symptoms items from the EORTC QLQ-C30 will be used to assess their severity, with the focus on assessments during the treatment period, and in the year following the end of treatment. These self-report instruments have been selected for this study due to the need for reliable and valid translations in multiple languages, given the international scope of this trial and the need to include a large number of participants.

Refer to Section 12.2.3 for patient reported outcomes hypotheses and objectives.

## 3.2.3 Study Population

Approximately 1800 patients with germline *BRCA* mutations (g*BRCA*m) and HER2 negative breast cancer who are at high risk of recurrence will be randomised into the trial.

All patients recruited in the study will be selected based on the following 3 principles:

- Genetic selection: Documented germline mutation in *BRCA1* or *BRCA2* that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function). Patients with germline *BRCA1* and/or germline *BRCA2* mutations that are considered to be non-detrimental (e.g. "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favour polymorphism" or "benign polymorphism," etc) will not be eligible for the study. In terms of *BRCA* mutation status, the following scenarios are considered:
  - Status known: for patients already known to have a gBRCA loss of function mutation (known as deleterious or suspected deleterious) the exact sequence variant must be recorded on the eCRF and a copy of the genetic diagnosis must be available at site. These patients may be randomised into the study based on the known status, however, re-confirmation of the loss of function mutation from a blood sample will be undertaken soon after randomisation by Myriad Genetic Inc.
  - Status unknown: The gBRCA mutation status must be determined by Myriad Genetic Inc. prior to randomisation as a loss of function mutation i.e. a known deleterious or suspected deleterious mutation
- **Phenotypic tumour selection:** All patients must have either TNBC or ER and/or PgR positive HER2 negative breast cancer as defined in the eligibility criteria section.
- **Prognostic factor selection:** Patients will be selected based on high risk of recurrence regardless of whether they received their chemotherapy in the adjuvant or neoadjuvant setting. High risk of recurrence will be defined as follows:
  - 1. For patients who underwent initial surgery and received adjuvant chemotherapy
    - TNBC patients must have been axillary node-positive (≥pN1, any tumour size) or axillary node negative (pN0) with invasive primary tumour pathological size > 2 cm (≥pT2)
    - ER and/or PgR positive/HER 2 negative patients must have had ≥4 pathologically confirmed positive lymph nodes.
  - 2. For patients who underwent neoadjuvant chemotherapy followed by surgery

- TNBC patients must have residual invasive breast cancer in the breast and/or resected lymph nodes (non pCR)
- ER and/or PgR positive/HER 2 negative patients must have residual invasive cancer in the breast and/or the resected lymph nodes (non pCR) AND a CPS&EG score ≥3. Instructions how to calculate CPS&EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix H.

#### 4. PATIENT SELECTION CRITERIA

Investigator(s) should keep a patient screening log of patients who entered pre-study screening.

Each patient should meet all of the inclusion criteria and none of the exclusion criteria for this study. Under no circumstances can there be exceptions to this rule.

Criteria relevant to Part 1 BRCA screening (Table 1) are marked with \*\* (double asterisk)

#### 4.1 Inclusion criteria

For inclusion in the study patients should fulfil the following criteria:

- 1. \*\*Provision of informed consent prior to any study specific procedures
- 2. \*\*Female or male patients must be  $\geq 18$  years of age
- 3A. For patients who underwent initial surgery and received adjuvant chemotherapy
  - TNBC patients must have been axillary node-positive (≥pN1, any tumour size) or axillary node-negative (pN0) with invasive primary tumour pathological size > 2 cm (≥pT2)
  - ER and/or PgR positive/HER 2 negative patients must have had ≥4 pathologically confirmed positive lymph nodes
- 3B. For patients who underwent neoadjuvant chemotherapy followed by surgery
  - TNBC patients must have residual invasive breast cancer in the breast and/or resected lymph nodes (non pCR)
  - ER and/or PgR positive/HER 2 negative patients must have residual invasive cancer in the breast and/or the resected lymph nodes (non pCR) AND a CPS&EG score ≥3. Instructions how to calculate CPS&EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix H

- 4. \*\*Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast that is one of the two following phenotypes:
  - a) TNBC defined as:
  - ER and PgR negative defined as IHC nuclear staining <1%.

#### **AND**

- HER2 negative (not eligible for anti-HER2 therapy) defined as:
  - o IHC 0, 1+ without ISH **OR**
  - o IHC 2+ and ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells **OR**
  - o ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells (without IHC)
- b) ER and/or PgR positive, HER2 negative breast cancer defined as:
- ER and/or PgR positive defined as IHC nuclear staining  $\geq 1\%$ .

#### AND

- HER2 negative (not eligible for anti-HER2 therapy) defined as:
  - IHC 0, 1+ without ISH **OR**
  - IHC 2+ and ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells OR</li>
  - ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells (without IHC)</li>

Patients with multifocal or multicentric invasive disease are eligible as long as all the lesions for which HER2 characterization is available are HER2 negative.

Patients with synchronous bilateral invasive disease are eligible as long as all the lesions assessed for HER2 on both sides are negative.

In both the above cases the lesion considered at highest risk for recurrence based on the investigator's discretion will be used for eligibility determination.

5. Documented germline mutation in *BRCA1* or *BRCA2* that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function)

Local *gBRCA* testing results, if available, will be used for establishing eligibility. If local *gBRCA* testing results are not available, central testing will be provided for those patients who otherwise appear to be eligible (see Section 6.2.1).

## 6A. Completed adequate breast surgery defined as:

- The inked margins of breast conservation surgery or mastectomy must be histologically free of invasive breast cancer and ductal carcinoma in situ with the exception of the posterior margin if this margin is the pectoralis major fascia or the anterior margin if this is the dermis. Patients with resection margins positive for lobular carcinoma *in situ* are eligible.
- Patients with breast conservation must have adjuvant radiotherapy. Patients
  having mastectomy may have adjuvant radiotherapy according to local policy
  and/or international guidelines.

#### 6B. Completed adequate axilla surgery defined as:

Adjuvant Chemotherapy Patients:

- Sentinel lymph node biopsy alone if negative or if lymph node(s) only contain micrometastases (≤2.0 mm) OR
- Positive sentinel lymph node biopsy followed by axillary nodal dissection or radiotherapy as per local guidelines OR
- Axillary dissection

Neoadjuvant Chemotherapy Patients:

- Sentinel lymph node biopsy performed *before* neoadjuvant chemotherapy:
  - If negative or if lymph node(s) only contain micrometastases
     (≤2.0 mm) additional axillary surgery is not required
  - If positive, axillary node dissection or axillary nodal radiotherapy should follow completion of neoadjuvant chemotherapy
- Sentinel lymph node biopsy performed *after* neoadjuvant chemotherapy:
  - If negative, additional axillary surgery not mandated

- If positive (micrometastases are regarded as positive), additional axillary surgery is required unless the patient is enrolled in a Phase III multicenter clinical trial proposing radiotherapy as alternative treatment of the axilla. The trial must be pre-approved by the OlympiA Executive Committee
- Axillary dissection
- 7. Completed at least 6 cycles of neoadjuvant or adjuvant chemotherapy containing anthracyclines, taxanes or the combination of both. Prior platinum as potentially curative treatment for prior cancer (e.g. ovarian) or as adjuvant or neoadjuvant treatment for breast cancer is allowed. (For neoadjuvant patients all chemotherapy should be delivered prior to surgery. No further cycles of chemotherapy post surgery are allowed.)
- 8. Patients must have adequate organ and bone marrow function measured within 28 days prior to randomisation with no blood transfusions (packed red blood cells and/or platelet transfusions) in the past 28 days prior to testing for organ and bone marrow function as defined below:
  - Haemoglobin ≥10.0 g/dL
  - Absolute neutrophil count (ANC)  $\geq 1.5 \times 10^9/L$
  - Platelet count  $\geq 100 \times 10^9/L$
  - Total Bilirubin ≤ ULN (institutional upper limit of normal) except elevated total bilirubin <1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin
  - AST (SGOT)/ALT (SGPT) ≤2.5 x ULN
  - ALP ≤2.5 x ULN

To rule out metastatic breast cancer, patients with screening ALT/AST or ALP above institutional upper limit of normal should have liver ultrasound, CT or MRI at any time point between diagnosis of current breast cancer and randomisation. Screening bone scan is required if ALP and/or corrected calcium level are above the institutional upper limit. (Note: PET CT scan may be used as an alternative imaging technique).

- 9. Serum or plasma creatinine  $\leq 1.5 \text{ x ULN}$
- 10. ECOG performance status 0-1

11A. Women who are not postmenopausal or have not undergone hysterectomy must have documented negative pregnancy test within 28 days prior to randomisation:

Postmenopausal is defined as:

- Age ≥60 years
- Age <60 years and amenorrheic for 1 year or more in the absence of chemotherapy and/or hormonal treatment
- Follicle stimulating hormone (FSH) and plasma estradiol levels in the postmenopausal range for women under 60 years
- Radiation-induced oophorectomy with last menses >1 year ago
- Bilateral oophorectomy
- \*\*Women of child bearing potential and their partners, who are sexually active, must agree to the use of two highly effective forms of contraception in combination. This should be started from the signing of the informed consent and continue, throughout the period of taking study treatment and for at least 1 month after last dose of study drug, or they must totally/truly abstain from any form of sexual intercourse. Male patients must use a condom during treatment and for 3 months after last dose of study drug when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception (see Appendix E for acceptable methods) if they are of childbearing potential.
- 12. \*\*Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
- 13. Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary tumour, mandatory\*.
  - \*NOTE: For adjuvant patients, this refers to the surgical specimen; for neoadjuvant patients, both the pre-treatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required.

14. Patient should be randomised in the trial ideally within a maximum of 8 weeks of completion of their last treatment (surgery, chemotherapy or radiotherapy), but in no case longer than 12 weeks.

#### 4.2 Exclusion criteria

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

- 1. \*\*Involvement in the planning and/or conduct of the study.
- 2. Patients who do not have deleterious or suspected deleterious *gBRCA1* and/or 2 mutations but only have *BRCA1* and/or *BRCA2* mutations that are considered to be non-detrimental (e.g., "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favour polymorphism" or "benign polymorphism" etc.).
- 3. \*\*Previous randomisation in the present study.
- 4. \*\*Evidence of metastatic breast cancer. Patient considered at high risk of having disseminated disease (i.e. those with locally advanced disease, clinical N2-3 or pathological N1-3 with the exception of pN1a in adjuvant patients) should have a CT/MRI scan of the Thorax/Abdomen/Pelvis or any other area as clinically indicated and a bone scan at any point between diagnosis of the current breast cancer and randomisation to rule out metastatic breast cancer. (Note PET/ CT scan may be used as an alternative imaging technique and precludes the need for bone scan). Patients with screening ALT/AST or ALP above institutional upper limit of normal should have liver ultrasound, CT or MRI at any time point between diagnosis of current breast cancer and randomisation. Screening bone scan is required if ALP and/or corrected calcium level are above the institutional upper limit. (Note PET/ CT scan may be used as an alternative imaging technique).
- 5. \*\*Exposure to an investigational product within 30 days or five half-lives (whichever is the longer) prior to randomisation.
- 6. \*\*Any previous treatment with a PARP inhibitor, including olaparib and/or known hypersensitivity to any of the excipients of study treatment.

- 7. \*\*Patients with second primary malignancy. **EXCEPTIONS** are:
  - o adequately treated non-melanoma skin cancer, curatively treated *in situ* cancer of the cervix, Ductal Carcinoma *in situ* (DCIS) of the breast, stage 1 grade 1 endometrial carcinoma.
  - other solid tumours and lymphomas (without bone marrow involvement) diagnosed ≥5 years prior to randomisation and treated with no evidence of disease recurrence and for whom no more than one line of chemotherapy was applied.
- 8. Resting ECG with QTc >470 msec detected on 2 or more time points within a 24-hour period or family history of long QT syndrome. If ECG demonstrates QTc >470 msec, patient will be eligible only if repeat ECG demonstrates QTc <470 msec.
- 9. Patients receiving systemic chemotherapy within 3 weeks prior to randomisation.
- 10. Patients receiving adjuvant radiotherapy within 2 weeks prior to randomisation.
- 11. Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks. Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
- 12. Persistent toxicities (≥CTCAE grade 2) caused by previous cancer therapy, excluding alopecia and CTCAE grade 2 peripheral neuropathy.
- 13. \*\*Patients with current or past history of haematologic malignancies and any clonal non-malignant haematological disorder which predisposes the patient to develop a haematological malignancy. Exception: lymphoma (refer to Exclusion Criterion 7).
- 14. Major surgery within 2 weeks prior to randomisation: patients must have recovered from any effects of any major surgery.

- 15. Patients considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
  - Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, extensive bilateral lung disease on High Resolution Computed Tomography scan or any psychiatric disorder that prohibits obtaining informed consent.
- 16. \*\*Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
- 17. Pregnant or breastfeeding women.
- 18. \*\*Patients with known active Hepatitis B or C or HIV
- 19. \*\*Previous allogeneic bone marrow transplant.
- 20. \*\*Whole blood transfusions in the last 120 days prior to entry to the study which may interfere with *gBRCA* testing (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no. 8)

For procedures for withdrawal of incorrectly enrolled patients see Section 5.3.

#### 5. STUDY CONDUCT

# 5.1 Restrictions during the study

# 5.1.1 Meals and dietary restrictions

It is prohibited to consume grapefruit juice while on study therapy.

#### 5.1.2 Contraception

Women of childbearing potential, who are sexually active, must agree to the use of two highly effective forms of contraception in combination (as described in Appendix E). This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug or they must totally/truly abstain from any form of sexual intercourse. Male patients must use a condom during treatment and for 3 months after last dose of study drug when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking olaparib and for 3 months following the last dose of olaparib. For details please refer to Appendix E Acceptable Birth Control Methods.
# 5.2 Patient enrolment and randomisation and initiation of study treatment

The following section outlines procedures for Screening Registration and for Randomisation, and for ordering Study Drug at randomisation:

- 1. The Investigator must obtain signed informed consent from the potential patient before any study specific procedures are performed.
- 2. The authorised site staff should register the patient for screening using the Frontier Science web-based Registration and Randomisation system. At the time of registration, the patient will be assigned a unique patient identifier (E-code) which should be used to identify the patient on the central Myriad sample, the eCRFs in Medidata Rave and any other trial-related communications.
- 3. The Investigator must determine patient eligibility. See Sections 4.1 and 4.2
- 4. If the patient meets the eligibility requirements, the authorised site staff should randomise the patient using the same Frontier Science web-based Registration and Randomisation system answering all questions which are asked by the system including questions relative to the stratification factors.
- 5. The randomisation system will randomly assign treatment (olaparib or placebo). The treatment allocation will be blinded for the Investigator and the patient.
- 6. Randomisation will automatically trigger initial study drug shipment to the site (except for countries where the initial drug shipment is sent upon site activation).
- 7. Once medication is received and confirmed in IVRS/IWRS, the site personnel can dispense the medication pack matching the kit identification number (Kit ID) assigned to the patient by the IVRS/IWRS drug ordering system.
- 8. Before dispensing, the site personnel should perform Kit verification transaction in IVRS/IWRS by matching the drug Kit ID with 2 letter security code printed on the medication pack's label.
- 9. Details of drug dispensing procedures can be found in the IVRS/IWRS manual.

## **5.2.1** Procedures for randomisation

Patient eligibility must be established before randomisation is undertaken. Randomisation can be performed for patients who met all eligibility criteria upon completion of all necessary Screening PART 2 procedures, either prior to or on Day 1, depending on the drug supply strategy for a particular country. This is to ensure that the study drug is available at site and can be dispensed to the patient during Visit 2 (Day1).

The randomisation system will use the following stratification factors:

- Hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC)
- NOTE: In cases of multifocal, multicentric or synchronous bilateral invasive disease, stratification is based on the status of the lesion considered at highest risk (at the investigator's discretion) that was used to determine eligibility.
- Neoadjuvant versus adjuvant chemotherapy
- Platinum therapy for current breast cancer: Yes/No

Eligible patients will be randomised in a 1:1 ratio to one of the following treatments:

- Olaparib tablets p.o. 300 mg twice daily
- Matching placebo tablets p.o. twice daily

It is recommended that patients commence study treatment within 7 days of randomisation, but no later than 21 days.

If, following randomisation, it is discovered that incorrect information on the stratification factors was entered at randomisation, then the correct information should be recorded in the eCRF but the randomisation system will retain the information that was provided at the time of randomisation

Further details about the randomisation process can be found in the Randomisation Guidelines

# 5.3 Procedures for handling patients incorrectly enrolled or randomised or initiated on study treatment

Patients who fail to meet the inclusion/exclusion criteria must not, under any circumstances, be enrolled or receive study medication. There can be no exceptions to this rule.

Where patients that do not meet the eligibility criteria are randomised in error or incorrectly started treatment, or where patients are subsequently found not to meet the pre-study criteria, a discussion should occur between the Study Physician or Medical Team (see Section 13.1) and the Investigator regarding whether to continue or discontinue the patient from treatment. Once a decision is made, Investigators need to ensure they comply with all applicable requirements for human patient protection and ethical review. The data on these patients will remain in the study database and will be included in appropriate analyses as defined by the Statistical Analysis Plan. Data values provided at the time of randomisation will not be changed. Any corrected values for stratification fields or other randomisation data fields will be recorded elsewhere in the clinical database, leaving the randomisation record to reflect the data actually provided at the time of randomisation.

Contact with the Study Physician or Medical Team (see Section 13.1) is to ensure all such decisions are appropriately documented. In situations where an agreement cannot be reached, the patient should have their study therapy stopped but should continue to have efficacy assessments as per the study plan, unless the patient withdraws consent.

## 5.4 Blinding and procedures for unblinding the study

#### 5.4.1 Methods for ensuring blinding

Olaparib and placebo treatment will be blinded.

The study medication will be labelled using a unique Kit ID number. The active and placebo tablets will be identical and presented in the same packaging to ensure blinding of the study medication.

# 5.4.2 Methods for unblinding individual patients

The treatment code for an individual patient should not be broken except in medical emergencies and when the appropriate management of the patient requires knowledge of the actual treatment assignment. The study investigator(s) can access unblinded patient information (i.e. randomised treatment information) through the IVRS/IWRS. The process for unblinding individual patients will be described in the IVRS/IWRS Manual that will be provided to each site. Following emergency unblinding the investigator should report the unblinding to the relevant Site Monitor, without revealing any treatment information.

Only life threatening situations should be considered as emergency such as in the cases listed below:

- Study drug was taken by someone else other than the patient by mistake.
- Patient is in a life threatening condition following intentional or unintentional consumption of study drug in higher doses than indicated.
- Patient admitted to emergency unit with what is regarded as life threatening condition irrespective of potential causal relationship with OLYMPIA study drug, and the treating team has to know the nature of all medications the patient is receiving.

Most other situations not mentioned above are regarded as non-emergency and hence the non-emergency unblinding procedure should apply.

Where a non-emergency unblinding is sought for an individual patient the process will require a discussion with the Study Physician or Medical Team (see Section 13.1) to understand the need for unblinding and help minimise any unnecessary unblinding, before the patient is unblinded. However the final decision as to whether or not to unblind the patient will be made by the investigator.

Disease progression or medical conditions that are manageable without any compromise to patient care in the absence of knowledge of the treatment received by the patient will not be considered as valid reasons for unblinding.

In both emergency and non-emergency cases, the information on the assigned treatment (i.e. Olaparib or Placebo) should be restricted only to the Principal Investigator and/or personnel involved in the clinical care of the patient as deemed appropriate by the Principal Investigator. This information should not be revealed to the sponsor or any member of the study team except for cases when the Monitor is required to access unblinded data to perform data verification in the eCRF.

Any patient unblinded by the site personnel will need to be immediately discontinued from the study treatment.

The AstraZeneca patient safety team retains the right to break the code for individual SAEs that are unexpected and are suspected to be causally related to the study treatment and that potentially require expedited reporting to regulatory authorities. Treatment codes will not be broken for the planned analyses of data until all decisions on the evaluability of the data from each individual patient have been made and documented and the target number of events has been reached.

#### 5.5 Treatments

#### 5.5.1 Identity of study treatment

AstraZeneca's Pharmaceutical Development, R&D Supply Chain will supply olaparib and matching placebo to the Investigator as green film-coated tablets as shown in Table 4 below.

Table 4 Identity of study treatment

| Study treatment | Dosage form and strength |
|---------------------------|---------------------------------|
| Olaparib* | Tablet −100 mg |
| Olaparib* | Tablet – 150 mg |
| Placebo to match olaparib | Tablet to match 100 mg olaparib |
| Placebo to match olaparib | Tablet to match 150 mg olaparib |

<sup>\*</sup> Descriptive information for olaparib can be found in the Investigator's Brochure

# 5.5.2 Doses and treatment regimens

## 5.5.2.1 Olaparib and matching placebo (study treatment)

Study treatment is available as a green film-coated tablet containing 150 mg or 100 mg of olaparib or matching placebo.

For all centres, olaparib and matching placebo (study treatment) will be packed in high-density polyethylene (HDPE) bottles with child-resistant closures. The randomised study

treatment will be dispensed to patients. Each dosing container will contain sufficient medication for at least each treatment period plus overage. The planned dose of 300 mg b.i.d. (twice daily) will be made up of two (2) x 150 mg tablets b.i.d. (twice daily) with 100 mg tablets used to manage dose reductions, as explained in Table 5.

Table 5 Study treatment doses and treatment regimens

| Total | Dose | Mor | ning | Evening | |
|---|---|---|---|---|---|
| daily dose | twice daily (b.i.d.) | Number of tablets | Tablet strength | Number of tablets | Tablet strength |
| 600 mg | 300 mg | 2 tablets | 150 mg | 2 tablets | 150 mg |
| Initial dose (3 | 00 mg twice daily | y) can be reduced | d as follows for A | AEs (no re-escala | tion allowed): |
| 500 mg | 250 mg | 1 tablet | 150 mg | 1 tablet | 150 mg |
| | | 1 tablet | 100 mg | 1 tablet | 100 mg |
| 400 mg | 200 mg | 2 tablets | 100 mg | 2 tablets | 100 mg |
| Temporary dose levels due to CYP3A inhibitor exposure (re-escalation allowed): | | | | | |
| 300 mg | 150 mg | 1 tablet | 150 mg | 1 tablet | 150 mg |
| 200 mg | 100 mg | 1 tablet | 100 mg | 1 tablet | 100 mg |

As soon as possible following randomisation, patients will be administered olaparib or matching placebo orally twice daily (b.i.d.) at 300 mg for 52 weeks. Two (2) x 150 mg olaparib or matching placebo tablets should be taken at the same time each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water. The olaparib/placebo tablets should be swallowed whole and not chewed, crushed, dissolved or divided. Olaparib/placebo tablets can be taken with a light meal/snack (e.g., two pieces of toast or two biscuits).

If vomiting occurs shortly after the study treatment tablets are swallowed, the dose should only be replaced if all of the intact tablets can be seen and counted. Should any patient enrolled on the study miss a scheduled dose for whatever reason (e.g., as a result of forgetting to take the tablets or vomiting), the patient will be allowed to take the scheduled dose up to a maximum of 2 hours after that scheduled dose time. If greater than 2 hours after the scheduled dose time, the missed dose is not to be taken and the patient should take their next allotted dose at the next scheduled time. Patient should not take two doses (4 tablets) at the same time.

Within this study, patients will not be provided olaparib post discontinuation of study treatment. Patients and investigators will not be routinely unblinded to study treatment prior to the final overall survival (OS) analysis.

#### 5.5.3 Additional study drug - Not applicable

## 5.5.4 Labelling

Labels will be prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfil GMP Annex 13 requirements for labelling. Label text will be translated into local language.

Specific dosing instructions will not be included on the label; the site must complete the "Patient Dispensing Card" with the details of the dosing instructions at the time of dispensing.

The patient emergency contact details will not be on the label, unless it is a country-specific regulatory requirement, but can be found in the informed consent and the 'Patient Dispensing Card'. For emergency purposes the patient must be in possession of the emergency contact details at all times.

# 5.5.5 Storage

All study drugs should be kept in a secure place under appropriate storage conditions. The study treatment label on the bottle specifies the appropriate storage.

### 5.5.6 Management of toxicity of study treatment

#### **General instructions**

- The CTCAE v4.0 must be used to grade the severity of AEs.
- All dose modifications should be based on the AE requiring the greatest modification.
- Therapy should be held until the AE returns to  $\leq$  grade 1 unless specified otherwise in the dose modification instructions.
- If study drug must be held for more than 4 weeks due to an AE or for any other reasons, permanently discontinue olaparib/placebo.
- Once a dose has been reduced, dose escalation is not permitted.
- If olaparib/placebo must be permanently discontinued, patient follow-up continues to be required as described in Table 2 and Table 3.
- If any other investigational treatment is administered, olaparib/placebo must be discontinued.

# 5.5.6.1 Study therapy following breast cancer recurrence or second primary cancer

Olaparib/placebo must be discontinued following diagnosis of breast cancer recurrence or diagnosis of a second primary malignancy (i.e., excluding new in situ carcinomas of any site and squamous or basal cell skin cancers). Further therapy is at the investigator's discretion.

## 5.5.6.2 Olaparib/placebo dose levels

All olaparib/placebo dose reductions are based on the dose levels listed in Table 6.

Any toxicity observed during the course of the study should be managed by guidelines as outlined in Table 7 Table 8 and Table 9. Once a dose has been reduced, dose re-escalation to a higher dose is not permitted.

Table 6 Olaparib/placebo dose levels

| | Dose Level (mg) twice daily | | | | |
|---|---|---|---|---|---|
| | Starting dose | Dose levels for AEs (no re-<br>escalation) | | Temporary do to CYP3A inhi exposure | |
| Olaparib/placebo | 300 | 250 | 200 | 150 | 100 |

Mandatory Treatment for Hematologic Toxicity and Treatment Guidance for other olaparib/placebo Toxicities Table 7

# Important table instructions:

| Dose modifications must be based on the AE requiring the greatest modification. | | | |
|---|---|---|---|
| | Adverse<br>Event | CTCAE<br>(v 4.0)<br>Grade | Action to be Taken |
| | Anaemia | 2<br>(8.0-9.5<br>g/dL) | Hold study therapy until > 9.5 g/dL: If recovery without packed red blood cells transfusion takes: 1-2 weeks – maintain dose; 3-4 weeks – ↓ one dose level If packed red blood cells transfusion given: reduce one dose level |
| Hematologic<br>Toxicity | | 3, 4 | Hold study therapy until > 9.5 g/dL:<br>$1^{st}$ appearance $-\downarrow 1$ dose level<br>$2^{nd}$ appearance $-\downarrow 2$ dose levels or discontinuation |
| Mandatory | Mandatory Neutrophil count decreased | 3 | Hold study therapy until ≥ 1200/mm <sup>3</sup> ↓ one dose level |
| (incl. febrile neutropenia) Platelet count decreased | (incl. febrile | 4 | Hold study therapy until ≥ 1200/mm <sup>3</sup> ↓ two dose levels |
| | 2 | Hold study therapy until ≥ 75,000//mm <sup>3</sup> $\downarrow$ one dose level | |
| | decreased | 3,4 | Hold study therapy until ≥ 75,000//mm <sup>3</sup> ↓ two dose levels |
| | Diarrhea (if | 2 | Maintain dose or ↓ one dose level |
| Other | attributable to olaparib/place | 3 | ↓ one dose level |
| toxicity<br>deemed to | bo) | 4 | Discontinuation |
| be | | 2 | Maintain dose or ↓ one dose level |
| attributable | attributable Mucositis – | 3 | ↓ one dose level |
| to study treatment | | 4 | Discontinuation |
| Guidance | Nausea (despite antiemetics) | 2 | Maintain dose or ↓ one dose level |
| | | 3 | ↓ one dose level |
| | | 2 | Maintain dose or ↓ one dose level |

### Important table instructions:

• Dose modifications must be based on the AE requiring the greatest modification.

| Dose modifications must be based on the AE requiring the greatest modification. | | | |
|---|---|---|---|
| | Adverse<br>Event | CTCAE<br>(v 4.0)<br>Grade | Action to be Taken |
| | Vomiting | 3 | ↓ one dose level |
| | (despite antiemetics) | 4 | ↓ one dose level or discontinuation |
| | Infection | 3 | Hold study therapy: When resolved: Maintain dose or ↓ one dose level Repeat appearance – ↓ one dose level |
| | | 4 | Hold study therapy: When resolved: ↓ two dose levels or discontinuation |
| Dyspnea | Dyspnea | 1, 2, 3 | Hold study therapy; rule out pneumonitis Follow instructions in footnote <sup>a</sup> |
| | | 4 | Discontinuation |
| | Pneumonitis | 2 | Follow instructions in footnote <sup>a</sup> |
| | Pneumonius | 3, 4 | Discontinuation |
| | Other | 2 | Maintain dose or ↓ one dose level |
| clinically significant AEs deemed related to study treatment b | 3 | ↓ one dose level | |
| | 4 | ↓ two dose levels or discontinuation | |

Hold olaparib/placebo and determine etiology. Unless prohibited based on instructions for other clinical diagnoses (i.e. other AEs), resume olaparib when grade 0 (if the AE requiring olaparib to be held was dyspnea) or when ≤ grade 1 (if the AE requiring olaparib to be held was ≥ grade 2).

Table 8 Dose reduction for study treatment to manage moderate renal impairment

| Initial dose | Moderate renal impairment (calculated creatinine clearance<br>by Cockcroft -Gault equation or based on a 24 hour urine<br>test between 31 and 50 ml/min): Dose reduction |
|---|---|
| 300 mg twice daily | 200 mg twice daily |

b Determination of "clinically significant" AEs is at the investigator's discretion.

Table 9 Dose reduction for study treatment with concurrent use of a strong or moderate CYP3A inhibitor

| Initial dose | Strong CYP3A inhibitor | Moderate CYP3A inhibitor |
|--------------------|------------------------|--------------------------|
| 300 mg twice daily | 100 mg twice daily | 150 mg twice daily |

For guidance on dose reductions for management of renal impairment refer to Section 5.5.6.3.

For guidance on dose reductions when concomitant strong or moderate CYP3A inhibitors cannot be avoided see section 5.6.2.

#### 5.5.6.3 Renal impairment

If subsequent to study entry and while still on study therapy, a patient's estimated creatinine clearance falls below the threshold for study inclusion (≥51 ml/min), retesting should be performed promptly.

A dose reduction is recommended for patients who develop moderate renal impairment (calculated creatinine clearance by Cockcroft-Gault equation or based on a 24 hour urine test of between 31 and 50 ml/min) for any reason during the course of the study: the dose of study treatment should be reduced to 200 mg b.i.d.

Because the creatinine clearance determination is only an estimate of renal function, in instances where the creatinine clearance falls between 31 and 50 mL/min, the investigator should use his or her discretion in determining whether a dose change or discontinuation of therapy is warranted.

Olaparib has not been studied in patients with severe renal impairment (creatinine clearance ≤30 ml/min) or end-stage renal disease; if patients develop severe impairment or end stage disease is it recommended that study treatment be discontinued.

### 5.5.6.4 Management of haematological toxicity

If blood transfusion support is required to maintain haemoglobin levels above 9.5 mg/dl at Dose Level -2 with no alternative explanation for the recurring anaemia, study treatment should be permanently discontinued and the patient referred for haematological evaluation.

If a patient develops febrile neutropenia, study treatment should be stopped and appropriate management including G-CSF may be given according to local hospital guidelines. If grade 3 or 4 anaemia, neutropenia or thrombocytopenia occurs, weekly differential blood counts including reticulocytes and peripheral blood smear should be performed until Hgb is > 9.5 mg/dl, ANC is  $> 1200/\text{mm}^3$  and platelets are  $> 75,000/\text{mm}^3$ . If persistent haematological toxicities lead to discontinuation of study therapy, the patient should be referred to a haematologist for further investigations. Differential blood counts including reticulocytes and

peripheral blood smear should be performed at least every 2 weeks until resolution or stabilization.

Bone marrow analysis and/or blood cytogenetic analysis should be considered at this stage according to standard haematological practice. Clinical notes and results from further testing should be submitted.

Development of a confirmed myelodysplastic syndrome or other clonal blood disorder should be reported as an SAE and full reports must be provided by the investigator to AstraZeneca Patient Safety.

Administration of blood cell products and platelet transfusions must be recorded in eCRF.

### 5.5.6.5 Management of new or worsening pulmonary symptoms

If new or worsening pulmonary symptoms (e.g., dyspnoea) or radiological abnormality occurs, study treatment should be held and a diagnostic workup (including a high resolution CT scan) should be performed, to exclude pneumonitis. Following investigation, if no evidence of abnormality is observed on CT imaging and symptoms resolve, then study treatment can be restarted, if deemed appropriate by the investigator. If significant pulmonary abnormalities are identified, these need to be discussed with the Study Physician or Medical Team (see Section 13.1).

## 5.5.6.6 Management of nausea and vomiting

No routine prophylactic anti-emetic treatment is required at the start of study treatment, however, patients should receive appropriate anti-emetic treatment at the first onset of nausea or vomiting and as required thereafter, in accordance with local treatment practice guidelines. As per international guidance on antiemetic use in cancer patients (ESMO, NCCN), generally a single agent antiemetic should be considered.

## 5.5.6.7 Interruptions for intercurrent non-toxicity related events

Study treatment dose interruption for conditions other than toxicity resolution should be kept as short as possible. If a patient cannot restart study treatment within 4 weeks for resolution of intercurrent conditions not related to disease recurrence or toxicity, the case should be discussed with AZ study physician. All dose reductions and interruptions (including any missed doses), and the reasons for the reductions/interruptions are to be recorded according to the eCRF guidelines. Study treatment should be stopped at least 3 days prior to planned surgery. After surgery study treatment can be restarted when the wound has healed. No stoppage of study treatment is required for any needle biopsy procedure. Study treatment should be discontinued for a minimum of 3 days before a patient undergoes radiation treatment. Study treatment should be restarted within 4 weeks as long as any bone marrow toxicity has recovered.

Because the AEs related to olaparib may include asthenia, fatigue and dizziness, patients should be advised to use caution while driving or using machinery if these symptoms occur.

# 5.6 Concomitant and subsequent treatment(s)

Any concomitant medications (exceptions described in Table 10) which are considered necessary for the patient's welfare, and which will not interfere with the study medication (in the opinion of the treating physician), may be given at the discretion of the investigator, providing the medications, the doses, dates and reasons for administration are recorded on the appropriate eCRF page in Medidata Rave.

Bisphosphonates or denosumab are allowed during study treatment phase and follow-up.

In addition, any relevant unplanned diagnostic, therapeutic or surgical procedure performed during the study period must be recorded. This includes any blood transfusions.

The reasons for the use, doses and dates of treatment should be recorded in the patient's medical records and appropriate sections of the eCRF.

All medications (prescriptions or over the counter medications) continued at the start of study or started during the study or until 30 days from the end of the last protocol treatment and different from the study medication must be documented.

Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse.

The receipt of other anti-neoplastic medications (with the exception of hormonal therapies as addressed in Section 5.6.1) and other investigational medication is prohibited during study treatment and follow-up.

Subsequent anti-cancer treatment is expected to be initiated following breast cancer recurrence; if subsequent anti-cancer treatment needs to be initiated during the 1-year treatment phase, study treatment must be stopped. Information on first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time must be recorded in the clinical database.

# 5.6.1 Administration of endocrine therapy

Patients should receive adjuvant endocrine therapy per local policy and/or international guidelines. Information on endocrine therapies should be collected and recorded in the eCRF until IDFS endpoint is met due to breast cancer related distant relapse.

# 5.6.2 Restricted concomitant medications

The use of any natural/herbal products or other traditional remedies should be discouraged but use of these products, as well as any medication or vaccine including over-the-counter or

prescription medicines, vitamins, and/or herbal supplements that the patient is receiving at the time of enrolment or receives during the study must be recorded along with:

- Reason for use
- Dates of administration including start and end dates

| Dosage information including dose and frequency Table 10 Restricted concomitant medications | |
|---|---|
| Medication/class of drug: | Usage (including limits for duration permitted and special situations in which it's allowed ): |
| Strong CYP3A inhibitors: itraconazole, telithromycin, clarithromycin, boosted protease inhibitors, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir | Strong or moderate CYP3A inhibitors should not be taken with study treatment. If there is no suitable alternative concomitant medication then the dose of study treatment should be reduced for the period of concomitant administration. The dose reduction of study treatment should be |
| Moderate CYP3A inhibitors: ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil | recorded in the CRF with the reason documented as concomitant CYP3A inhibitor use. |
| | • Strong CYP3A inhibitors – reduce the dose of study treatment to 100 mg b.i.d for the duration of concomitant therapy with the strong inhibitor and for 5 half-lives afterwards. |
| | <ul> <li>Moderate CYP3A inhibitors - reduce the<br/>dose of study treatment to 150 mg b.i.d for<br/>the duration of concomitant therapy with<br/>the moderate inhibitor and for 3 half-lives<br/>afterwards.</li> </ul> |
| | <ul> <li>After the washout of the inhibitor is<br/>complete, the study treatment dose can be<br/>re-escalated.</li> </ul> |
| Strong CYP3A inducers: | Strong or moderate CYP3A inducers should not be taken with study treatment. |
| phenobarbital, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine, enzalutamide and St John's Wort | If the use of any strong or moderate CYP3A inducers are considered necessary for the patient's safety and welfare this could diminish |
| Moderate CYP3A inducers: | the clinical efficacy of olaparib. If a patient requires use of a strong or moderate |

Moderate CYP3A inducers: bosentan, efavirenz and modafinil

If a patient requires use of a strong or moderate CYP3A inducer then they must be monitored carefully for any change in efficacy of study treatment.

Table 10 Restricted concomitant medications

| Medication/class of drug: | Usage (including limits for duration permitted and special situations in which it's allowed ): |
|---|---|
| <ul> <li>CYP3A4 substrates: hormonal contraceptive, simvastatin, cisapride, cyclosporine, ergot alkaloids, fentanyl, pimozide, sirolimus, tacrolimus and quetiapine</li> <li>CYP2B6 substrates: bupropion, efavirenz</li> <li>OATP1B1substrates: bosentan, glibenclamide, repaglinide, statins and valsartan</li> <li>OCT1, MATE1 and MATE2K substrates: metformin</li> <li>OCT2 substrates: serum creatinine</li> <li>OAT3 substrates: furosemide, methotrexate</li> </ul> | Effect of olaparib on other drugs Based on limited in vitro data, olaparib may increase the exposure to substrates of CYP3A4, OATP1B1, OCT1, OCT2, OAT3, MATE1 and MATE2K. Based on limited in vitro data, olaparib may reduce the exposure to substrates of 2B6. Caution should be observed if substrates of these isoenzymes or transporter proteins are co-administered. |
| Anticoagulant therapy | Patients who are taking warfarin may participate in this trial; however, it is recommended that international normalised ratio (INR) be monitored carefully at least once per week for the first month, then monthly if the INR is stable. Subcutaneous heparin and low molecular weight heparin are permitted. |
| Administration of other anti-cancer agents | Patients must not receive any other concurrent anti-cancer therapy, including investigational agents, while on study treatment. Patients may continue the use of bisphosphonates or denosumab. |

#### 5.6.3 Anti-emetics/Anti-diarrheals

Should a patient develop nausea, vomiting and/or diarrhoea, then these symptoms should be reported as AEs (see Section 6.4.3) and appropriate treatment given.

### 5.6.4 Live virus and bacterial vaccines

Live virus and bacterial vaccines should not be administered whilst the patient is receiving study treatment and during the 30-day follow-up period. An increased risk of infection by the administration of live virus and bacterial vaccines has been observed with conventional chemotherapy drugs and the effects with olaparib are unknown.

# 5.7 Treatment compliance

The administration of all study drugs during the 1-year treatment phase of the study should be recorded in the appropriate sections of the eCRF.

Patients should be given clear instructions on how and when to take their study treatment. Patients will self-administer study treatment. Study site staff should do a tablet count at regular intervals during treatment. Compliance will be assessed by the tablet count and the information should be recorded in the appropriate section of the eCRF. After the tablet count has been performed, the remaining tablets will not be returned to the patient, but will be retained by the investigative site until reconciliation is completed by the study monitor. All patients must return their bottle(s) of study treatment at the appropriate scheduled visit, when a new bottle will be dispensed. Patients should be instructed to notify study site personnel of missed doses. Site staff will then complete the relevant eCRF pages to document the drug actually given.

Patients should return all containers at the next scheduled visit and any remaining tablets at the End of Treatment visit.

#### 5.7.1 Accountability

The study drug provided for this study will be used only as directed in the study protocol.

The study personnel will account for all study drugs dispensed to and returned from the patient.

Study site personnel will account for all study drugs received at the site, unused study drugs and for appropriate destruction. Certificates of delivery, destruction and return should be signed and retained. Any discrepancies must be accounted for on the appropriate forms.

## 5.8 Discontinuation of study treatment

Patients may be discontinued from the study treatment in the following situations:

- Patient decision. The patient is free at any time to discontinue study treatment, without prejudice to further clinical care
- Adverse Event
- Completion of 12 months treatment period
- Confirmed pregnancy during treatment
- Severe non-compliance with study protocol

- Loco-regional breast cancer recurrence (ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence)
- Distant breast cancer recurrence
- Contralateral invasive breast cancer or second primary non-breast invasive cancer
- Death
- Bone marrow findings consistent with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML)

## 5.8.1 Procedures for discontinuation of a patient from study treatment

A patient that decides to discontinue study treatment should always be asked about the reason(s) and the presence of any adverse events. If possible, he/she will be seen and assessed by an investigator(s). Adverse events will be followed up (See Sections 6.4.3 and 6.4.4); questionnaires and all study drugs should be returned by the patient.

If a patient is withdrawn from study, see Section 5.9.

If patients discontinue study treatment early, the site monitor must be informed immediately.

Any patient discontinuing prior to completing 52 weeks of study treatment should attend the treatment discontinuation visit, if possible. Thereafter the patient should be seen at 30 days post discontinuation for the evaluations outlined in the study schedule.

After premature discontinuation of study treatment, the principal investigator/sub-investigator will continue to provide appropriate clinical care and, as far as possible, follow the study visit schedule. Only the visits where efficacy assessments are scheduled should be performed i.e. week 12, 24, 38, 52 (as applicable) in Year 1 and all visits in Year 2 onwards. Only the following assessments should be done: recurrent/new cancers assessment, mammogram and/or breast MRI, and Quality of Life questionnaires.

Collection of vital signs, AEs, haematology/clinical chemistry results and concomitant medications is no longer required. Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse. The date of discontinuation, the reasons, and details of the following specific cancer therapies (first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time) should also be recorded on the eCRF.

Samples should be collected at disease recurrence per protocol: blood biomarker samples (mandatory) and tumour sample (optional). If a recurrent/new cancer assessment is scheduled

within 4 weeks of the study treatment discontinuation visit, it can be performed at the 30 day follow-up visit.

Patients who meet the IDFS endpoint while on study therapy should attend the treatment discontinuation visit and follow up visit 30 days after the last dose of study treatment. See Section 3 for guidelines on subsequent study visits, which are dependent on which IDFS endpoint has been met.

After discontinuation of study treatment at any points in the study, all ongoing AEs or SAEs must be followed until resolution unless, in the investigator's opinion the condition is unlikely to resolve due to the patients underlying disease, or the patient is lost to follow-up (see Sections 6.4.3 and 6.4.4). All new AEs and SAEs occurring during the 30 calendar days after the last dose of study medication must be reported (if SAEs, they must be reported to AstraZeneca via both the eCRF and paper SAE report to AstraZeneca data entry site (DES) within 24 hours as described in Section 6.4.4) and followed to resolution as above. Patients should be seen at least 30 days after discontinuing study medication to collect and / or complete AE information.

# 5.9 Withdrawal from study

Patients are at any time free to withdraw from study (study treatment and assessments), without prejudice to further clinical care (withdrawal of consent). Such patients should always be asked about the reason(s) and the presence of any adverse events. If possible, they will be seen and assessed by an investigator. Adverse events will be followed up (See Sections 6.4.3 and 6.4.4); questionnaires (e.g. for patient reported outcomes) and all study drugs should be returned by the patient.

Withdrawn patients will not be replaced.

Reasons for withdrawal from the study:

- Voluntary withdrawal by the patient who is at any time free to discontinue their participation in the study, without prejudice to further treatment\*
- Incorrectly enrolled patients i.e., the patient does not meet the required inclusion/exclusion criteria for the study this option is only applicable to patients not randomised into the study (i.e. screen failures identified prior to randomisation)
- Patient lost to follow-up
- Death

<sup>\*</sup> If a patient decides at any point in the trial that they do not wish to continue with the full study schedule of assessments but are still willing to provide important study information (e.g. disease recurrence information and/or survival status information) then the patient should

continue in the study and information should continue to be collected in the eCRF. However if a patient does not wish to have any further data collected, only then should they be considered as withdrawing consent from the study. To minimise the number of cases of early withdrawal the investigator should discuss the options with the patient to see if they would still be willing to provide information on the important study endpoints (disease recurrence and overall survival), in which case they would remain in the study.

If a patient withdraws consent (i.e. no further assessment or collection of their data) he/she should be specifically asked if they are also withdrawing consent to the use of any of their samples (tumour and blood) taken during the trial (see Section 6.6, 6.7 and 6.8).

Data obtained prior to withdrawal of consent will be maintained in the clinical database and used in the study reporting.

#### 6. COLLECTION OF STUDY VARIABLES

## 6.1 Recording of data

A Web Based Data Capture (WBDC) Medidata Rave system will be used for data collection and query handling. This system is provided by Frontier Science. The investigator will ensure that data are recorded on the eCRFs as specified in the study protocol and in accordance with the instructions provided.

The investigator will sign the completed eCRFs when requested by the Frontier Science Data Management Team. A copy of the completed eCRFs will be archived at the study site.

## 6.2 Study procedures

A study initiation visit must be conducted at the centre prior to the commencement of any study activities requiring informed consent. A schedule for the tests and evaluations to be conducted in this study is contained in this section and in Table 1, Table 2 and Table 3.

### **6.2.1** Screening procedures

The following assessments, procedures and data collection should be performed during screening as per Figure 1 and Table 1:

- Provision of informed consent
- Assessment of eligibility against inclusion/exclusion criteria
- Date of birth
- Current and concomitant medications including previous cancer therapies
- Medical and surgical history including previous cancer and radiotherapy and history of blood transfusions in previous 120 days

- Family history of cancer
- Physical examination
- Vital signs (blood pressure and pulse; body temperature), body weight, height
- ECG (within 28 days prior to randomisation)
- Haematology/Clinical chemistry/Coagulation (see Section 6.4.5.2)/Urinalysis
- ECOG Performance Status
- If a patient with conservative surgery does not have a mammogram or breast MRI within 12 months prior to Screening PART 1, then this assessment must be performed prior to randomisation. Breast imaging should be performed on any remaining intact breast. Radiological tests to exclude a second primary breast cancer (either ipsilateral and/or contralateral) are mandatory before enrolment (within 12 months prior to Screening PART 1) for patients with any remaining intact breast tissue (including male patients). The preferred tests are mammograms or MRI (MRI preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion.
- Pregnancy tests on serum or urine samples will be performed for women of childbearing potential within 28 days prior to randomisation on Day 1 of the study prior to commencing treatment.
- CPS+EG score (Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS)) for the non-pCR patients who received prior neoadjuvant chemotherapy (Mittendorf et al 2011; Jeruss et al 2008). Instructions on how to calculate the CPS&EG score are provided in Appendix H.
- Patient Reported Outcomes and Quality of life questionnaire: FACIT-Fatigue and EORTC QLQ-C30 will be collected prior to randomisation once eligibility is confirmed.
- Germline BRCA 1/2 mutation status determination
  - All patients must have a known deleterious or suspected deleterious germline BRCA mutation to be randomised; this may have been determined by local genetic testing prior to enrolment into the study or may be assessed as part of the enrolment procedure for the study which requires a central laboratory test at Myriad Genetics Inc.

- Two blood samples are mandated for all patients, one sample will be used to test for *BRCA* mutations using the current commercial Myriad BRCAnalysis test, and the second sample is required for a bridging study to validate the companion diagnostic test for olaparib.
- O Patients with unknown *BRCA* status must have a central test performed by Myriad prior to randomisation into the study. Patients will need to have met the locally agreed guidelines for *BRCA* testing with genetic counselling arranged as appropriate. When the result from the Myriad test indicates the patient does have a deleterious or suspected deleterious *BRCA* mutation, and the patient meets all other eligibility criteria, the patient can be randomised into the study. Specimen collection and results disclosure to the potential subject will be conducted using local ethical procedures.
- o It is recommended that, where required, the Myriad gBRCA test is undertaken during adjuvant or neoadjuvant chemotherapy to allow time for necessary counselling and for the return and discussion of the test result.
- O Patients with known deleterious or suspected deleterious *BRCA* mutation/s prior to enrolment into the study can be randomised into the study based on this local result provided they meet all other eligibility criteria. The specific *BRCA1/2* mutation must be reported in the clinical database by selecting the appropriate value from the drop down menu. At screening, reconfirmation of the *BRCA* mutation from a blood sample will be undertaken by a central laboratory (Myriad Genetic Inc). Should the result from the central Myriad test indicate that the patient does not have a deleterious or suspected deleterious *BRCA* mutation, this information will be available to the study investigator and the decision as to whether or not the patient continues study treatment should be made between the patient and study investigator.
- o If the discordance is based on the absence of the alteration identified in the local laboratory by the central laboratory, then analysis of a second specimen, collected independently from the patient and sent to Myriad Genetics for reanalysis of the presence or absence of the mutation specified in the original test or otherwise as discussed with Myriad laboratory staff, may be performed under the protocol, to eliminate sample mislabelling and similar errors. These errors are expected to be uncommon. If the discordance is based on interpretation of the pathogenicity of an alteration identified by both laboratories (i.e., Myriad classifies the alteration as neither deleterious nor suspected deleterious), a repeat test will not be indicated. The OlympiA trial Genetic Advisory Committee can be consulted if needed.

See Section 6.6.2 for gBRCA Myriad samples collection.

- Adverse events must be captured from time of main consent. Any medical condition (new or worsening of a pre-existing condition) that occurs post Screening PART 2 and is continuing at randomisation should be recorded in Medical History in the eCRF as a medical condition current at randomisation. If the condition worsens post randomisation, this should be recorded as an AE/SAE in the eCRF with start date as the date the grade worsened and the new grade should be reported on the AE form. The AE/SAE would be considered to have resolved when it resolves to the baseline grade, not to zero. Any medical condition considered of clinical relevance (new or worsening of a pre-existing condition) that occurs post consent for PART 2 and resolves prior to randomisation should also be recorded as medical history. In Screening PART 1 of the study only SAEs related to study mandated procedures (i.e. blood draw) will be collected and reported to AstraZeneca DES via the paper SAE report. In Screening PART 2 all SAEs will be collected and reported via the paper SAE report to AstraZeneca DES within 24 hours. For the patients who experienced an SAE in either Screening PART 1 or PART 2 that were eventually randomised, the SAE should be reported in the eCRF retrospectively in addition to paper reporting as described in Section 6.4.4.
- Check availability of an archival paraffin embedded tumour tissue sample (see Section 6.6.3). (The sample will only be submitted to the study bio-repository once the patient has been randomised)
- Check availability of an archival paraffin embedded post neoadjuvant tumour tissue sample (see Section 6.6.4). (The sample is required from neoadjuvant patients only and will only be sent to the study bio-repository once the patient has been randomised)

The Principal Investigator/Sub-Investigator should adhere to the study plan, procedures and perform tests/observations in accordance with the protocol.

#### **6.2.2** On-treatment assessments

Patients will attend the clinic on day 1 (1st day of treatment) and, following the commencement of 300 mg b.i.d. twice daily dosing, every 2 weeks during the first month, every 4 weeks for the following 5 months and 3 monthly for the remaining 6 months of study treatment plus 30 days after its discontinuation.

The following assessments will be performed at time points specified in the study schedule (see Section 3.1, Table 1 and Table 2):

Physical examination (data does not need to be entered in the eCRF, however any clinically significant changes from baseline must be reported as an AE or an event)
 e.g. any signs of recurrence of disease should be reported

- ECOG performance status: if assessed within 7 days of randomisation, it should not be assessed again at day 1 of study treatment
- Vital signs (blood pressure and pulse rate, body temperature, body weight): if assessed within 7 days of randomisation, are not required to be assessed again at day 1 of 1st day of study treatment
- Haematology and clinical chemistry: Safety blood samples do not need to be repeated on Day 1 of study treatment if there have been separate assessments within 7 days before randomisation and at least 3 weeks after last dose of chemotherapy, unless the investigator believes that it is likely to have changed significantly
- Race and ethnicity unless collection of this data is not allowed by local regulations
- Pregnancy tests on serum or urine samples will be performed for women of childbearing potential. If the test is positive the patient is ineligible/must be discontinued from study treatment immediately.
- AE and concomitant medications (including any blood transfusions) at every visit
- Patient Reported Outcomes and Quality of life questionnaire: FACIT-Fatigue and EORTC QLQ-C30 will be collected at 6 months, 12 months, 18 months and 24 months



- Optional pharmacokinetic samples will be obtained from consenting patients on day 29 (see Section 6.8)
- Optional tumour biopsy at disease recurrence (Section 6.6.5)
- Mandatory blood sample for biomarker analysis (e.g. cfDNA) on day 1 prior to first dose of study treatment, 30 days post study treatment and disease recurrence (Section 6.6.6)
- Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory during study participation (starting at week 24 and yearly thereafter) for patients with any remaining intact breast tissue (including male patients). The preferred tests are mammogram or MRI (MRI preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and

radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion.

#### Dispensing of and return of unused study treatment

Within this study, patients will not be provided olaparib post discontinuation of study treatment. Patients and investigators will not be unblinded to study treatment prior to the final overall survival (OS) analysis.

### 6.2.3 Efficacy follow-up assessments

Assessments for disease recurrence, new cancers and overall survival will be performed based on signs and symptoms, clinical assessment (i.e. physical exam), mammograms and/or breast MRI and vital status

Following randomisation, during the first 2 years patients will be assessed for disease recurrence and new cancers every 3 months. During years 3, 4 and 5 patients will be assessed every 6 months and then annually until approximately 10 years from randomisation if an IDFS endpoint due to a distant breast cancer relapse has not been met.

Mammograms and/or MRI (MRI preferred for patients younger than 50 years) (ipsilateral and/or contralateral) will be performed annually in patients with retained breast tissue beginning 6 months after first day of treatment for approximately 10 years if an IDFS endpoint due to a distant breast cancer relapse has not been met.

Once a patient has received clinical follow-up for efficacy for approximately 10 years, or an IDFS endpoint due to a distant breast cancer relapse has been met, the patient will then enter the annual survival follow-up phase of the study. During the survival follow-up phase, no clinic visits will be required; information may be collected via telephone, medical records or death registries. Vital status information, as well as other information specified in footnote g of Table 2 will be collected until 10 years after the last patient is randomised.

In addition to disease status and vital status, information on first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time, including those received during the survival follow-up phase, will be collected. Information on endocrine therapies should be collected and recorded in the eCRF until IDFS endpoint is met due to breast cancer related distant relapse. The therapy type and start and stop dates of therapy will be collected.

# 6.2.4 Safety follow-up assessments 30 days after last dose of olaparib/placebo

A follow-up visit should be conducted 30 days after the last dose of olaparib/placebo. Any serious and/or non-serious AEs ongoing at the time of discontinuation of study treatment or which have occurred during the defined 30-day follow-up period must be followed up (in accordance with Section 6.4.3). Appropriate safety evaluations should be repeated and/or

additional tests performed at any time when clinically indicated, or at the discretion of the investigator, until resolution, unless, in the investigator's opinion, the condition is unlikely to resolve due to the patient's underlying disease. If the patient is lost to follow-up, then this should be noted in the eCRF. The assessments to be carried out at the 30-day follow-up visit are detailed in the study schedule (Table 2).

See Section 6.4.3 for details of long term safety collection.

## 6.2.5 Patient management post-primary analysis

The data cut off (DCO) for the primary analysis for IDFS will occur once 330 IDFS events have been reported. Once this data is fully validated the primary analysis will be conducted and reported.

At the time of the DCO for the primary analysis patients will continue in the study as per the protocol following the outlined study plan assessments. Patients who have completed treatment and all relevant safety assessments will continue to have regular efficacy assessments as detailed in the study plan. All ongoing patients will continue to be followed for recurrence, new cancers and overall survival irrespective of treatment status.

It is anticipated that further analysis of the efficacy data, particularly the secondary endpoints, will be conducted with more mature follow-up. Any further available safety data will also be reported.

### 6.2.6 Patient management post-final analysis

Study follow-up will continue until approximately 10 years after the last patient is randomised. After this time no further data collection is anticipated.

Patient management post the final analysis will be according to local clinical practice. All patients will have completed study treatment by the time of the final analysis.

#### 6.3 Efficacy

#### **6.3.1** Tumour evaluation

All treatment decisions and analysis for this study will be based on investigator evaluation of assessments. Following randomisation, all patients will be assessed regularly for signs, symptoms and evidence of disease recurrence by reviewing medical history, performing physical examination and mammogram and/or breast MRI (MRI preferred for patients younger than 50 years) see Table 2 and Table 3. Efficacy assessments (medical history and physical examination) will be performed on a 3 monthly basis during the first 2 years, followed by 6 monthly assessments for years 3, 4 and 5 and annually thereafter. All patients will have mammogram and/or breast MRI (ipsilateral and/or contralateral) annually for approximately 10 years beginning 6 months after day 1. Evidence of disease recurrence or new primary cancer will require histopathological and/or radiological confirmation.

Patients will be regularly assessed, through clinical visits, for recurrence (local and distant) and new cancers for approximately 10 years follow-up regardless of whether they have discontinued study treatment or started any subsequent anti-cancer therapies. Following completion of approximately 10 years' clinical follow-up assessments, patients will enter a survival follow-up phase, which will continue until 10 years after the last patient is randomised. During the survival contact period information on any known subsequent sites of metastases, new cancers and further subsequent therapies (information on first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time) will be captured as well as vital status. Study visits are not required during the survival follow-up phases; contact will be made via telephone, medical records or death registries once per year.

Loco-regional recurrence of the disease (ipsilateral or regional invasive breast cancer) should be cytologically/histologically confirmed. Imaging to assess for distant metastatic disease or any other area as clinically indicated should be performed at the time of local recurrence to ensure that any further spread of the disease is detected. Isolated loco-regional recurrence should be managed with curative intent when possible. Suspected distant recurrence should be confirmed by radiological examination and every attempt be made to obtain histopathological confirmation when a metastatic lesion is easily accessible for biopsy. Invasive contralateral breast cancer or invasive non-breast secondary primary cancer should be confirmed by histopathology.

Patients who develop loco-regional recurrence should discontinue study treatment (if within the study treatment period) but will continue to be followed for distant recurrence (including subsequent sites of metastases) and all new cancers (local, regional, second primary malignancy or contralateral breast cancer), subsequent therapies and survival as per study schedule. The first EVENT (local, regional or distant recurrence, second primary malignancy or contralateral breast cancer) should be recorded in the eCRF. The following additional information should also be recorded in the eCRF along with results of confirmatory tests:

- First distant relapse (if not the first EVENT);
- CNS metastases, that should always be reported regardless of any prior recurrences;
- Loco-regional relapses, occurring after the first event;
- Contralateral breast cancer, at any time;
- Any second primary malignancies, at any time.

Patients who develop distant recurrence should discontinue study treatment (if within the study treatment period) but will continue to be followed for development of additional sites of metastatic disease, new cancers, subsequent therapies and survival as per the survival follow-up schedule.

Disease recurrence or new cancers should be reported in the eCRF as soon as possible after they are discovered. This includes events diagnosed during study visits but also any event diagnosed during non-study visits.

Once known, death information should also be recorded in the eCRF as soon as possible.

## 6.4 Safety

The Principal Investigator is responsible for ensuring that all staff involved in the study is familiar with the content of this section.

## 6.4.1 Definition of adverse event (AE)

An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g. nausea, chest pain), signs (e.g. tachycardia, enlarged liver) or the abnormal results of an investigation (e.g. laboratory findings, electrocardiogram).

The term AE is used to include both serious and non-serious AEs.

## 6.4.2 Definitions of serious adverse event (SAE)

A serious adverse event is an AE occurring during any study phase (i.e. from the time a patient signs a study specific consent form, treatment, and follow-up), that fulfils one or more of the following criteria:

- Results in death
- Is immediately life-threatening
- Requires in-patient hospitalisation or prolongation of existing hospitalisation
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital abnormality or birth defect
- Is an important medical event that may jeopardise the patient or may require medical intervention to prevent one of the outcomes listed above.

For further guidance on the definition of an SAE, see Appendix A to the Clinical Study Protocol.

## 6.4.3 Recording of adverse events

#### Time period for collection of adverse events

Adverse events will be collected from time of signature of main informed consent\* throughout the treatment period up to and including the 30-day follow-up period. All ongoing and any new AEs/SAEs identified during the 30 calendar days follow-up period after the last dose of study medication must be followed to resolution unless the event is considered by the investigator to be unlikely to resolve, or the patient is lost to follow-up or in survival follow-up. AstraZeneca retains the right to request additional information for any patient with ongoing AE(s)/SAE(s) at the end of the study, if judged necessary. Any medical condition (new or worsening of a pre-existing condition) that occurs post Screening PART 2 and is continuing at randomisation should be recorded in medical history in the eCRF as a medical condition current at randomisation. If the condition worsens post randomisation, this should be recorded as an AE/SAE in the eCRF with start date as the date the grade worsened and the new grade should be reported on the AE form. The AE/SAE would be considered to have resolved when it resolves to the baseline grade, not to zero. Any medical condition considered of clinical relevance (new or worsening of a pre-existing condition) that occurs post consent for PART 2 and resolves prior to randomisation should also be recorded as medical history. Any AE happening from randomisation to the 30-day follow-up period should be reported on the AE form in the eCRF. If an Investigator learns of any SAEs, including death, at any time after a patient has completed 30 days post treatment follow-up period, and he/she considers there is a reasonable possibility that the event is causally related to the study treatment, the investigator should notify AstraZeneca, Patient Safety by reporting the SAE via both the eCRF in Medidata Rave and paper SAE report to AstraZeneca DES.

Any case of MDS/AML or new primary malignancy occurring at any time from signature of informed consent for the entire participation of the patient in the study including the follow-up period should be reported as an SAE. Non-melanoma skin cancers need to be reported as a non-serious AE unless at least one of the seriousness criteria is met and then it must be reported as an SAE, see Section 6.4.2. Any of these types of serious or non-serious events need to be reported to AstraZeneca Patient Safety according to SAE reporting procedures for this study, regardless of investigator's assessment of causality or knowledge of the treatment arm. If a patient develops MDS/AML, full diagnostic details and classification should be provided e.g. bone marrow and cytogenetic analysis reports, see Sections 5.5.6.3 and 6.4.5.5. A questionnaire will be sent to any investigator reporting MDS/AML or new primary malignancy so that relevant details can be reported.

\*In Screening PART 1 of the study only SAEs related to study mandated procedures (i.e. blood draw) will be collected and reported to AstraZeneca DES via the paper SAE report. In Screening PART 2 all SAEs will be collected and reported via the paper SAE report to AstraZeneca DES within 24 hours. For the patients who experienced an SAE in either Screening PART 1 or PART 2 that were eventually randomised, the SAE should be reported in the eCRF retrospectively in addition to paper reporting as described in Section 6.4.4.

# Adverse events after the 30 day follow up period

For pharmacovigilance purposes and characterisation, any SAE of MDS/AML, new primary malignancy, or pneumonitis occurring after the 30 day follow up period should be reported to AstraZeneca Patient Safety regardless of investigator's assessment of causality or knowledge of the treatment arm. After all follow up visits investigators should report the occurrence of any MDS/AML or any new primary malignancies as per protocol.

At any time after a patient has completed the study, if an investigator learns of any SAE including sudden death of unknown cause, and he/she considers there is a reasonable possibility that the event is causally related to the investigational product, the investigator should notify AstraZeneca, Patient Safety.

Otherwise, after study treatment completion (i.e. after any scheduled post treatment follow-up period has ended) there is no obligation to actively report information on new AEs or SAEs occurring in study patients. This includes new AEs/SAEs in patients still being followed up for survival but who have completed the post treatment follow up period (30 days).

#### Follow-up of unresolved adverse events

Any SAE or non-serious adverse event that is still ongoing during the 30-day follow-up visit must be followed up to resolution unless the event is considered by the investigator to be unlikely to resolve, or the patient is lost to follow-up. AstraZeneca may request additional information for any patient with ongoing AE(s)/SAE(s) at the end of the study, if necessary.

#### Variables

The following variables will be collected for each AE;

- AE description (verbatim)
- The dates when the AE started and stopped
- CTCAE grade and changes in CTCAE grade
- Whether the AE is serious or not
- Investigator causality rating against the study treatment (yes or no)
- Action taken with regard to study treatment
- Outcome.

In addition, the following variables will be collected for SAEs:

Date that the AE met criteria for serious AE

- Date Investigator became aware of serious AE
- Reason for AE being considered serious
- Date of hospitalisation
- Date of discharge
- Probable cause of death
- Date of death
- Autopsy performed
- Causality assessment in relation to Study treatment or procedure(s)
- Causality assessment in relation to Other medication
- Description of AE.

## **Severity of AE**

For each episode of an adverse event, all changes to the CTCAE grade attained as well as the highest attained CTC grade should be reported.

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria in Section 6.4.2. An AE of severe intensity should not necessarily be considered serious. For example, nausea that persists for several hours may be considered severe nausea, but not an SAE. On the other hand, a stroke that results in only a limited degree of disability may be considered a mild stroke but would be an SAE.

The grading scales found in the National Cancer Institute (NCI) CTCAE version 4.0 will be utilised for all events with an assigned CTCAE grading. For those events which do not fall under any of the CTCAE defined categories, the investigator should assess them as mild, moderate, severe, or life-threatening, or, if the patient dies, as an event leading to the patient's death.

A copy of the CTCAE version 4.0 can be downloaded from the NCI Cancer Therapy Evaluation Program website http://ctep.cancer.gov/.

#### **Causality collection**

The Investigator will assess causal relationship between study treatment and each Adverse Event, and answer 'yes' or 'no' to the question 'Do you consider that there is a reasonable possibility that the event may have been caused by the study treatment?'

For SAEs causal relationship will also be assessed for other medication and study procedures. Note that for SAEs that could be associated with any study procedure the causal relationship is implied as 'yes'.

A guide to the interpretation of the causality question is found in Appendix A to the Clinical Study Protocol.

#### Adverse events based on signs and symptoms

All AEs spontaneously reported by the patient or reported in response to the open question from the study personnel: 'Have you had any health problems since the previous visit/you were last asked?', or revealed by observation will be collected and recorded in the eCRF. When collecting AEs, the recording of diagnoses is preferred (when possible) rather than recording a list of signs and symptoms. However, if a diagnosis is known and there are other signs or symptoms that are not generally part of the diagnosis, the diagnosis and each sign or symptom will be recorded separately.

#### Adverse events based on examinations and tests

The reporting of laboratory/vital signs/ECG abnormality as an AE should be avoided unless one of the following is met:

- Any criterion for an SAE is fulfilled
- Causes study treatment discontinuation
- Causes study treatment interruption
- Causes study treatment dose reduction
- The investigator believes that the abnormality should be reported as an AE

If deterioration in a laboratory value/vital sign is associated with clinical signs and symptoms, the sign or symptom will be reported as an AE and the associated laboratory result/vital sign will be considered as additional information. Wherever possible the reporting investigator uses the clinical, rather than the laboratory term (e.g. anaemia versus low haemoglobin value). In the absence of clinical signs or symptoms, clinically relevant deteriorations in non-mandated parameters should be reported as AE(s).

Deterioration of a laboratory value, which is unequivocally due to disease recurrence, should not be reported as an AE/SAE.

Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the baseline assessment will be reported as an AE.

**NB.** Cases where a patient shows an AST or ALT  $\ge 3x$ ULN or total bilirubin  $\ge 2x$ ULN may need to be reported as SAEs, please refer to Appendix D 'Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law', for further instructions.

#### Disease recurrence

The development of loco-regional recurrence or distant metastasis to the primary cancer under study should be considered as disease progression and not an AE. Events, which are unequivocally due to disease recurrence, should not be reported as an AE during the study.

#### New cancers

The development of a new primary cancer should be reported as an AE (see Section Olaparib adverse events of special interest) and would in most cases meet seriousness criteria (with the exception of some non-melanoma skin cancers). New primary cancers are those that are not the primary reason for the administration of the study treatment and have developed after the inclusion of the patient into the study. They do not include metastases of the original cancer. Symptoms of metastasis or the metastasis itself should not be reported as an AE/SAE, as they are considered to be disease recurrence. New primary cancers are considered as IDFS event and must also be reported on the endpoint CRF. Patients with new primary cancers that can be adequately treated with surgery only and which do not require any additional (neo)adjuvant treatment of any kind can continue to receive investigational product and be followed for secondary endpoints. Rules regarding temporary interruption due to surgery apply (see Section 5.5.6.7). Patients with new primary cancers which require (neo)adjuvant treatment of any kind for appropriate management must be discontinued from study treatment.

#### Deaths

All deaths that occur during the study must be reported as follows:

- Death that is clearly the result of breast cancer recurrence or progression should be reported to the study monitor at the next monitoring visit and should be documented in the DEATH eCRF but should not be reported as an SAE.
- Where death is not due (or not clearly due) to breast cancer recurrence or progression of the disease under study, the cause of death must be reported to the study monitor as an SAE within 24 hours (see Section 6.4.4 for further details). The report should contain a comment regarding the co-involvement of progression of disease, if appropriate, and should assign main and contributory causes of death. This information should be captured in the relevant eCRF.

Deaths with an unknown cause should always be reported as an SAE. A post mortem maybe helpful in the assessment of the cause of death, and if performed a copy of the post-mortem results should be forwarded to AstraZeneca Patient Safety within the usual timeframes.

## Olaparib adverse events of special interest

Adverse events of special interest (AESI) are events of scientific and medical interest specific to the further understanding of olaparib's safety profile and require close monitoring and rapid communication by the investigators to AstraZeneca. Adverse Events of Special Interest for olaparib are MDS/AML, new primary malignancy (other than MDS/AML) and pneumonitis.

A questionnaire will be sent to any investigator reporting an AESI by AstraZeneca Patient Safety, as an aid to provide further detailed information on the event. During the study there may be other events identified as AESIs that require the use of a questionnaire to help characterise the event and gain a better understanding regarding the relationship between the event and study treatment.

## 6.4.4 Reporting of serious adverse events

All SAEs have to be reported, whether or not considered causally related to the study treatment, or to the study procedure(s). All SAEs will be recorded in the eCRF and AstraZeneca Patient Safety Database.

If any SAE occurs in the course of the study, then investigators or other site personnel should inform their site monitor immediately, or **no later than 24 hours** after being made aware of it.

The designated study representative works with the investigator to ensure that all the necessary information is provided to the AstraZeneca Patient Safety data entry site via the paper SAE report and is completed in the eCRF within one calendar day of initial receipt for fatal and life threatening events and within five calendar days of initial receipt for all other SAEs.

For fatal or life-threatening adverse events where important or relevant information is missing, active follow-up is undertaken immediately. Investigators or other site personnel inform the site monitor of any follow-up information on a previously reported SAE immediately, or **no later than 24 hours** after being made aware of it.

If the WBDC system is not available, then the Investigator or other study site personnel reports an SAE to the appropriate AstraZeneca representative via the paper SAE report and while eCRF is completed immediately upon its availability.

The AstraZeneca representative will advise the Investigator/study site personnel how to proceed.

## 6.4.5 Laboratory safety assessment

Blood and urine samples for determination of clinical chemistry, haematology, coagulation, and urinalysis will be taken at the times indicated in the Study Schedule (see Table 1 and Table 2).

These tests will be performed by the hospital's local laboratory. Additional analyses may be performed if clinically indicated.

Any clinically significant abnormal laboratory values should be repeated as clinically indicated and recorded on the eCRF.

The following laboratory variables will be measured:

## 6.4.5.1 Full haematology assessments for safety

- haemoglobin
- red blood cells [RBC]
- platelets
- mean cell volume [MCV]
- mean cell haemoglobin concentration [MCHC]
- mean cell haemoglobin [MCH]
- white blood cells [WBC]
- absolute differential white cell count
  - (neutrophils, lymphocytes, monocytes, eosinophils and basophils) and absolute neutrophil count or segmented neutrophil count and Band forms should be performed at each visit and when clinically indicated. If absolute differentials not available please provide % differentials

### 6.4.5.2 Coagulation

- activated partial thromboplastin time (APTT) will be performed at baseline and if clinically indicated
- international normalised ratio (INR) will be performed at baseline and if clinically indicated unless the patient is receiving warfarin. Patients taking warfarin may participate in this study; however, it is recommended that prothrombin time (INR and APTT) be monitored carefully at least once per week for the first month, then monthly if the INR is stable

## 6.4.5.3 Clinical chemistry assessments for safety

- sodium
- potassium

- calcium
- creatinine
- total bilirubin
- alkaline phosphatase [ALP]
- aspartate transaminase [AST]
- alanine transaminase [ALT]
- urea or blood urea nitrogen [BUN]
- total protein
- albumin

**NB.** If a patient has AST **or** ALT ≥3xULN **or** total bilirubin ≥2xULN please refer to Appendix D "Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law", for further instructions.

For blood volume see Section 7.1.

#### 6.4.5.4 Urinalysis

Urinalysis by dipstick should be performed at baseline and then only if clinically indicated. Microscopic analysis should be performed by the hospital's local laboratory if required.

### 6.4.5.5 Bone marrow or blood cytogenetic samples

Bone marrow or blood cytogenetic samples may be collected for patients with prolonged haematological toxicities as defined in Section 5.5.6.3.

Bone marrow analysis should include an aspirate for cellular morphology, cytogenetic analysis and flow cytometry, and a core biopsy for bone marrow cellularity. If it is not possible to conduct cytogenetic analysis or flow cytometry on the bone marrow aspirate, then attempts should be made to carry out the tests on a blood sample. Full reports must be provided by the investigator for documentation on the Patient Safety database.

### 6.4.6 Physical examination

For timing of individual measurement refer to study schedule (Table 1, Table 2 and Table 3). A physical examination will be performed according to site's local practice.

Clinical signs and symptoms of disease recurrence should be further investigated as appropriate (please refer to Section 6.3).

#### **6.4.7 ECG**

## 6.4.7.1 Resting 12-lead ECG

ECGs are required during screening within 28 days prior to randomisation.

Twelve-lead ECGs will be obtained after the patient has been rested in a supine position for at least 5 minutes. The investigator or designated physician will review the paper copies of each of the timed 12-lead ECGs.

ECGs will be recorded at 25 mm/sec. All ECGs should be assessed by the investigator as to whether they are clinically significantly abnormal / not clinically significantly abnormal. If there is a clinically significant abnormal finding, the investigator will record it as an AE on the eCRF. The original ECG traces must be stored in the patient medical record as source data.

### 6.4.8 Vital signs

Height will be assessed at screening only.

Weight will be assessed at screening and as clinically indicated at any other time.

Any changes in vital signs should be recorded as an AE, if applicable.

The date of collection and measurement will be recorded on the appropriate eCRF.

#### 6.4.8.1 Pulse and blood pressure

Blood pressure and pulse rate will be measured preferably using a semi-automatic BP recording device with an appropriate cuff size. For timings of assessments refer to the Study Schedule (see Table 1 and Table 2).

The date of collection and measurement will be recorded on the appropriate eCRF.

### **6.4.8.2** Body temperature

Body temperature will be measured in degrees Celsius at the times indicated in the Study Schedule (see Table 1 and Table 2).

The date of collection and measurement will be recorded on the appropriate eCRF.

## 6.4.9 Other safety assessments

#### 6.4.9.1 Serum or urine pregnancy test

Pregnancy tests on serum or urine samples will be performed for women of childbearing potential within 28 days prior to randomisation (Table 1), on Day 1 of the study prior to commencing treatment, at the time points shown in Table 2 during study treatment and at the 30 day follow up visit. Tests will be performed by the hospital's local laboratory. If results are

positive the patient is ineligible/must be discontinued from study treatment immediately. Details of the pregnancy tests must be recorded in the patient's medical records.

## 6.5 Patient reported outcomes (PRO)

## 6.5.1 FACIT-Fatigue

The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F Scale) is a 13-item questionnaire that assesses patient self-reported fatigue and its impact upon daily activities and function (Yellen et al 1997). Response options for each item range from 0 (Not at all) to 4 (Very much), where higher scores indicate greater patient-reported fatigue. The FACIT-F scale was originally developed to evaluate fatigue associated with anaemia in cancer patients and has been used as an endpoint in clinical trials in various cancer populations including breast cancer and non-small cell lung cancer. Content validity of the FACIT-F has been demonstrated in a large sample of mixed cancer patients (n>300). Reliability (internal consistency, test-retest reliability, criterion validity, and responsiveness/sensitivity to change) of the FACT-F has also been documented (Yellen et al 1997).

## 6.5.2 EORTC QLQ-C30

In this study patient-reported disease related symptoms and health-related quality of life (HRQoL) will be evaluated using the validated EORTC QLQ-C30 questionnaire (Aaronson et al 1993). The EORTC QLQ-C30 questionnaire was developed to assess HRQoL and is the most commonly used cancer-specific tool in oncology. It has undergone extensive testing and validation as well as detailed cross-cultural testing and validation and has been used in breast cancer trials.

The EORTC QLQ-C30 comprises 30 questions designed for all cancer types. Questions can be grouped into the following subscales:

- 5 multi-item functional scales (physical, role, emotional, cognitive and social functioning)
- A 2-item global health status scale
- Symptom scales/items
  - 3 multi-item symptom scales (fatigue, pain, nausea and vomiting)
  - Dyspnoea
  - Insomnia
  - Appetite loss
  - Constipation
- Diarrhoea
- Financial difficulties

# 6.5.3 Administration of PRO questionnaires

FACIT-Fatigue and EORTC QLQ-C30 questionnaires will be collected at baseline (within screening period after eligibility confirmed but prior to randomisation) and then 6 months, (24 weeks), 12 months (52 weeks), 18 months and 24 months following randomisation.

Questionnaires shall be administered to a patient by delegated site personnel (e.g., a research nurse, study coordinator) adequately trained and listed on Site's Delegation Log. Site shall assign a trained back-up person to cover if that individual is absent. The AZ Study Delivery Team (or delegate) will provide relevant training in administration of the questionnaires. The significance and relevance of the data need to be explained carefully to participating patients so that they are motivated to comply with data collection.

The instructions for completion of the PRO questionnaires are as follows:

- They must be completed at the clinical visit prior to any other study procedures (following informed consent) and before discussion of disease progress to avoid biasing the patient's responses to the questions. They must be completed in private by the patient
- The patient should be given sufficient time to complete at their own speed
- The patient should not receive help from relatives, friends or clinic staff to answer the questionnaire. However, if the patient is unable to read the questionnaires (e.g., is blind or illiterate) the questionnaires may be read out by trained clinic staff and responses recorded
- On completion of the questionnaires they should be handed back to the person responsible for questionnaires who should check for completeness
- Only one answer should be recorded for each question.

The site staff should enter the information directly into the eCRF.

After the baseline, questionnaires are to be administered at follow-up visits, so that when a follow-up visit is delayed, completion of the questionnaire may also be delayed. Patients who experience disease recurrence or diagnosis of a second primary cancer will not be expected to continue with the PRO assessments. Patients who discontinue study drug for other reasons will be expected to continue the PRO assessments per protocol schedule. Patients who never initiate study medication should not continue to complete PRO assessments. If a patient declines to complete a scheduled PRO assessment or if the questionnaire is not completed for

any other reason (and cannot be completed by phone or mail), a Quality of Life Missing Data eCRF page should be completed by the institution instead.

#### 6.6 Biomarkers

Tumour and blood samples will be collected for mandated and optional biomarker work as detailed in the Laboratory Manual.

For blood volume see Section 7.1

#### 6.6.1 Biomarker samples

The archival diagnostic tumour sample is mandated\* and the screening blood samples for *BRCA* mutation status are mandated.

Table 11 Samples for Biomarker Research

| Sample Type | Visits | <b>Optional or Mandatory</b> |
|---|---|---|
| Whole blood sample for prospective germline <i>BRCA</i> testing at central laboratory for patients with unknown <i>BRCA</i> status and for confirmation of <i>BRCA</i> status for those with previous results | Screening | Mandatory |
| Whole blood sample for assessment of current and future <i>BRCA</i> mutation assay(s) | Screening | Mandatory |
| Archival tumour sample | | |
| Surgical tumour samples for adjuvant patients | Screening | Mandatory* for all randomised patients |
| Pre-treatment diagnostic core biopsy for neoadjuvant patients | Screening | Required* for all randomised patients |
| Surgical tumour sample post neoadjuvant chemotherapy | Screening | Required* for all randomised neoadjuvant patients |
| On-study disease recurrence tumour biopsy | At disease recurrence | Optional |
| Blood samples (plasma and serum) for biomarker analysis | Day 1 prior to first<br>dose of study<br>treatment, 30 days<br>post study treatment<br>discontinuation,<br>disease recurrence | Mandatory |

<sup>\*</sup> For adjuvant patients, this refers to the surgical specimen; for neoadjuvant patients, both the pretreatment core biopsy and the surgical specimen with residual disease are requested but only one is

mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required.

The samples and data from this research will be coded and not identified with any personal details. Each sample will be identified with the study and patient enrolment number. In this way biomarker data may be correlated with clinical data, samples destroyed in the event of withdrawal of consent and regulatory audit enabled. However, only the investigator will be able to link the biomarker sample to the individual patient. Research biomarker data may be generated in real time during the study or retrospectively and will have unknown clinical significance. The study investigative team will not provide research biomarker results to patients, their family members, any insurance company, an employer, clinical study investigator, general physician or any other third party unless required to do so by law. The patient's samples will not be used for any purpose other than those described in the protocol.

The gBRCA status result from the Myriad assessment for patients with unknown BRCA status will be provided to the investigator and will be collected as part of the patient's demography and medical history details.

#### 6.6.2 Collection of blood sample for Myriad germline BRCA1 and BRCA2 testing

Two blood samples are mandated for all patients. One sample will be used to test for *BRCA* mutations using the current commercial Myriad BRCAnalysis test. This result will confirm or determine subject eligibility. The second sample is required for a bridging study to validate the companion diagnostic test for olaparib (see Section 6.6.2.1 below).

All patients must have a known deleterious or suspected deleterious germline *BRCA* mutation to be randomised; this may have been determined by local genetic testing prior to study entry or may be assessed as part of the enrolment procedure for the study (via central testing by Myriad), see Section 6.2.1. The specific g*BRCA* alteration on which eligibility is based must be entered into the trial database by selecting the appropriate value from the drop down menu. If the central laboratory analysis does not confirm a local g*BRCA* determination, that information should also be entered in the eCRF, along with an indication of whether or not the patient was enrolled into the trial.

Residual blood (or its derivatives) may be used to evaluate future BRCA companion diagnostic tests and for additional exploratory work, to elucidate the mechanism of response, understand the mode of action of study treatment, and improve the understanding of disease recurrence (including BRCA mutation status and its role in response).

For blood volume see Section 7.1.

# 6.6.2.1 Collection of a blood sample for assessment of current and future *BRCA* mutation assay(s)

At the time that the sample is collected for shipment to Myriad for central testing, all patients will be required to provide a second mandatory 9 ml blood sample that will be stored for subsequent assessment of current and future *BRCA* mutation assay(s).

Samples may also be used to investigate future BRCA mutation assays as well as mutations in other genes known/predicted to have a role in breast cancer.







# 6.8 Pharmacokinetics (optional)

PK sampling (optional) will be performed in a subset of patients. Each patient participating in this component of the study will be asked to provide 5 blood samples, one from each of the pre-defined time windows below, preferably on visit 4, day 29. Nevertheless, the samples can also be taken at a later treatment visit, provided that PK consent was obtained beforehand.

- Pre-dose (before morning dose)
- Between 0 and 0.5 hour post-dose
- Between >0.5 and 1.5 hour post-dose
- Between 3 and 6 hours post-dose
- Between >6 and 12 hours post-dose (before evening dose)

# 6.8.1 Pharmacokinetic samples (Subset of patients)

Approximately 150 patients randomised to olaparib/placebo, at pre-agreed sites will have PK assessment samples taken.

#### 6.8.2 Collection of samples

PK samples are to be taken as a blood sample (2 mL) for determination of olaparib concentrations in plasma. It is essential that PK blood sampling is conducted within the protocol sample collection windows indicated above.

To ensure that the assessments are carried out in the correct order, and that PK sampling is conducted within the required sampling window, it will be necessary to arrange the assessment procedures so that the PK assessments fall on/around the correct timing (see Section 6.8). The actual time of dosing and collection of all PK samples must be recorded as described below:

It is essential that the time of collection of all 5 PK samples is recorded and that the times of the morning and evening dose on the day of PK sampling and the time of dose the evening before is recorded.

Samples will be collected, labelled, stored and shipped as detailed in the Laboratory Manual.

For blood volume see Section 7.1.

#### 6.8.3 Determination of drug concentration

Samples for determination of olaparib concentrations in plasma will be analysed by Covance on behalf of Clinical Bioanalysis Alliance, AstraZeneca R&D, using an appropriate bioanalytical method. Full details of the analytical method used will be described in a separate bioanalytical report. Placebo samples will not be analysed unless specified.

Full instructions for collection, labeling, storage and shipment of samples are provided in the Laboratory Manual. Results will only be reported for samples shipped within a timeframe for which the stability of olaparib in the samples has been validated and shown to be acceptable.

#### 6.9 Health economics

# 6.9.1 Resource use (serious adverse events)

Resource use for serious adverse events (including hospitalisations) will be captured through the adverse reporting procedures described in Section 6.4.

#### 7. BIOLOGICAL SAMPLING PROCEDURES

# 7.1 Volume of blood

The volume of blood that will be drawn from each patient will vary, depending upon the length of time that the patient remains in the trial and if the patient is in the subset of patients having PK samples taken. However, the total volume of blood to be drawn from each patient in the study (including for PK samples), assuming they complete screening, 12 months of treatment, a treatment discontinuation visit and the 30-day follow-up visit, should not exceed 208 mL.

Safety laboratory assessments will be performed locally at each centre's laboratory by means of their established methods. The number of samples/blood volumes is therefore subject to site-specific change.

Extra blood samples may also be collected if, for example, additional samples are required for repeat safety assessments or *BRCA* testing.

The total volume of blood that will be drawn from each patient in this study is as follows:

Table 12 Volume of blood to be drawn from each patient

| Assessment | | Sample volume (mL) | No. of samples | Total volume<br>(mL) |
|---|---|---|---|---|
| Safety | Clinical chemistry | 5 | 13 | 65 |
| | Haematology | 5 | 13 | 65 |
| | Coagulation | 5 | 1 | 5 |
| Whole blood sample for Myriad <i>BRCA</i> test (retrospective/prospective) | | 9 | 1 | 9 |
| Whole blood sample for assessment of current and future <i>BRCA</i> mutation assay(s) | | 9 | 1 | 9 |
| | | 1 | | |
| Serum Pregnancy test | | Site dependent | Site may use urine instead | |
| | | ı | I | I |
| | | 1 | I | I |
| | | J | | |
| | | | | • |
| | | • | • | • |
| | | I | I | |
| Pharmacokinetic (<br>processed to plasr | (Blood samples<br>ma & frozen) (Optional) | 2 | 5 | 10 |
| Total | | | | 208 |

# 7.2 Handling, storage and destruction of biological samples

The samples may be used up, disposed of after analyses or retained for further use as described here.

Biological samples for future research will be retained at the study bio-repository for a maximum of 15 years following the Last Patient's Last Visit in the study. The results from future analysis will not be reported in the Clinical Study Report but separately in a Scientific Report.

Biosamples collected for this study will be stored in study specific bio-repositories that are under the guardianship of BIG (non-US samples) and NRG Oncology and NCI (US samples) on behalf of the study Steering Committee.

## 7.2.1 Pharmacogenetic samples

The processes adopted for ensuring confidentiality of samples for genetic analysis are important. Samples will be stored for a maximum of 15 years, from the date of the Last Patient's Last Visit, after which they will be destroyed. DNA is a finite resource that may be used up during analyses. Samples will be stored and used until no further analyses are possible or the maximum storage time has been reached after which samples will be destroyed.

DNA will be extracted from the blood sample. The DNA sample will be assigned a unique number replacing the information on the sample tube. Thereafter, the DNA sample will be identifiable by the unique DNA number only. The DNA number is used to identify the sample and corresponding data at the AstraZeneca genetics laboratories, or at the designated contract laboratory. No personal details identifying the individual will be available to any person (AstraZeneca employee or contract laboratory staff working with the DNA.)

The samples and data for genetic analysis in this study will be single coded. The link between the patient enrolment/randomisation code and the DNA number will be maintained and stored in a secure environment, with restricted access within the Clinical Genotyping Group Laboratory Information Management System (LIMS) at AstraZeneca. The link will be used to identify the relevant DNA samples for analysis, facilitate correlation of genotypic results with clinical data, allow regulatory audit and to trace samples for destruction in the case of withdrawal of consent when the patient has requested disposal/destruction of collected samples not yet analysed.

#### 7.2.2 Pharmacokinetic samples

Pharmacokinetic samples will be disposed of after the Bioanalytical Report finalisation or six months after issuance of the draft Bioanalytical Report (whichever is earlier), unless required for future analyses. Additional analyses may be conducted on the anonymised, pooled pharmacokinetic samples to further evaluate and validate the analytical method. Any results from such analyses will be reported separately from the Clinical Study Report (CSR).

Sample reproducibility analysis, if any, will be performed alongside the bioanalysis of the test samples. The results from the evaluation will not be reported in the CSR but separately in a Bioanalytical Report. Anonymised samples will be retained for no longer that 12 months after the Bioanalytical Report is finalised.

# 7.3 Labeling and shipment of biohazard samples

The Principal Investigator should ensure that samples are labelled and shipped in accordance with the Laboratory Manual and the Biological Substance, Category B Regulations (materials containing or suspected to contain infectious substances that do not meet Category A criteria), see Appendix B 'IATA 6.2 Guidance Document'.

Any samples identified as Infectious Category A materials should not be shipped and no further samples will be taken from the patient unless agreed with AstraZeneca/BIG or Partners and appropriate labelling, shipment and containment provisions are approved.

#### 7.4 Chain of custody of biological samples

A full chain of custody is maintained for all samples throughout their lifecycle.

The Principal Investigator at each centre is responsible for ensuring full traceability of collected biological samples from the patients while in storage at the centre until shipment or disposal (where appropriate).

The sample receiver keeps full traceability of the samples while in storage and during use until used or disposed of or until further shipment and keeps documentation of receipt of arrival.

AstraZeneca/BIG/NRG Oncology and their Partners keep oversight of the entire life cycle through internal procedures, monitoring of study sites and auditing of external laboratory providers.

Biosamples collected for this study will be stored in study specific bio-repositories that are under the guardianship of BIG (non-US samples) and NRG Oncology and NCI (US samples) on behalf of the study Steering Committee.

Samples retained for further use are registered in the bio-repositories systems during the entire sample life cycle.

If required, the remaining biological samples are returned to the site, according to local regulations or at the end of the retention period, whichever is the sooner.

# 7.5 Withdrawal of informed consent for donated biological samples

If a patient withdraws consent to the use of donated biological samples, the samples will be disposed of/destroyed, and the action documented. If samples are already analysed,

AstraZeneca/BIG/NRG Oncology and their Partners are not obliged to destroy the results of this research.

*BRCA* sample: As collection of the biological samples is an integral part of the study, then the patient is withdrawn from further study participation.

Archival tumour sample: Although mandatory\*, the patient may continue in the study if the patient is already randomised.

\* For adjuvant patients, this refers to the surgical specimen; for neoadjuvant patients, both the pre-treatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and reembedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required.

Tumour samples at relapse: As collection of the biological samples is an optional part of the study, then the patient may continue in the study.

Pharmacokinetic samples: As collection of the pharmacokinetic samples is an optional part of the study, then the patient may continue in the study.

Blood samples for biomarker analysis (e.g. cfDNA): Collection of the biological samples is a mandatory part of the study, however, the patient may continue in the study despite withdrawing consent for analysis of the biomarker samples.

Blood sample for pharmacogenetic analysis: As collection of the biological samples is an optional part of the study, then the patient may continue in the study.

The Principal Investigator/site staff:

- Should ensure that the Site Monitor is notified immediately of a patient's withdrawal of informed consent for the use of donated samples
- Should ensure that biological samples from that patient, if stored at the study site, are immediately identified, disposed of /destroyed, and the action documented
- Should ensure that the laboratory(ies) holding the samples is/are informed about the withdrawn consent immediately and that samples are disposed/destroyed, the action documented and the signed document returned to the study site

• Should ensure that the patient and Site Monitor are informed about the sample disposal.

The Site Monitor ensures that the central laboratory(ies) holding the samples is/are informed about the withdrawn consent immediately and that samples are disposed of/destroyed and the action documented and returned to the study site.

# 8. ETHICAL AND REGULATORY REQUIREMENTS

#### 8.1 Ethical conduct of the study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/Good Clinical Practice, applicable regulatory requirements and the AstraZeneca policy on Bioethics and Human Biological Samples.

# 8.2 Patient data protection

The Informed Consent Form will incorporate (or, in some cases, be accompanied by a separate document incorporating) wording that complies with relevant data protection and privacy legislation.

AstraZeneca will not provide individual genotype results to patients, any insurance company, any employer, their family members, general physician or any other third party, unless required to do so by law.

Extra precautions are taken to preserve confidentiality and prevent genetic data being linked to the identity of the patient. In exceptional circumstances, however, certain individuals might see both the genetic data and the personal identifiers of a patient. For example, in the case of a medical emergency, a study medical representative or an investigator might know a patient's identity and also have access to his or her genetic data. Also Regulatory authorities may require access to the relevant files, though the patient's medical information and the genetic files would remain physically separate.

The exception to the above is the result of the Myriad gBRCA test. This will be made available to the Investigator and patient.

# 8.3 Ethics and regulatory review

An Institutional Review Board (IRB)/Ethics Committee should approve the final study protocol, including the final version of the Informed Consent Form and any other written information and/or materials to be provided to the patients. The investigator will ensure the distribution of these documents to the applicable Ethics Committee, and to the study site staff.

The opinion of the Ethics Committee should be given in writing. The investigator should submit the written approval to AstraZeneca/BIG/Partners (and the CTSU for US centres) before enrolment of any patient into the study.

The Ethics Committee should approve all advertising used to recruit patients for the study.

AstraZeneca/BIG/Partners (and NRG Oncology/CTEP for US centres) should approve major modifications to the Informed Consent Form that are needed to meet local requirements.

If required by local regulations, the protocol should be re-approved by the Ethics Committee annually.

Before enrolment of any patient into the study, the final study protocol, including the final version of the Informed Consent Form must be approved by the national regulatory authority or a notification to the national regulatory authority must be done, according to local regulations.

AstraZeneca/BIG/Partners will handle the distribution of these documents to the national regulatory authorities.

AstraZeneca/BIG/Partners will provide Regulatory Authorities, Ethics Committees and Principal Investigators with safety updates/reports according to local requirements, including SUSARs (Suspected Unexpected Serious Adverse Reactions), where relevant.

Each Principal Investigator is responsible for providing the Ethics Committees/IRB with reports of any serious and unexpected adverse drug reactions from any other study conducted with the investigational product. AstraZeneca will provide this information to the Principal Investigator so that he/she can meet these reporting requirements.

#### 8.4 Informed consent

The Principal Investigator(s) at each centre will:

- Ensure each patient is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study
- Ensure each patient is notified that they are free to discontinue from the study at any time
- Ensure that each patient is given the opportunity to ask questions and allowed time to consider the information provided
- Ensure each patient provides signed and dated informed consent before conducting any procedure specifically for the study
- Ensure the original, signed Informed Consent Form(s) is/are stored in the Investigator's Study File
- Ensure a copy of the signed Informed Consent Form is given to the patient

• Ensure that any incentives for patients who participate in the study as well as any provisions for patients harmed as a consequence of study participation are described in the informed consent form that is approved by an Ethics Committee.

### 8.5 Changes to the protocol and informed consent form

Study procedures will not be changed without the mutual agreement of the International coordinating Investigator, National Co-ordinating Investigator, and the Principal Investigator and AstraZeneca/BIG/NRG Oncology/Partners and the study Steering Committee.

If there are any substantial changes to the study protocol, then these changes will be documented in a study protocol amendment and where required in a new version of the study protocol (Revised Clinical Study Protocol).

Any protocol amendment must be approved by the relevant Ethics Committee and if applicable, should obtain the national regulatory authority approval, before implementation. Local requirements are to be followed for amended protocols.

AstraZeneca will distribute any subsequent amendments and new versions of the protocol to each Principal Investigator(s). For distribution to Ethics Committee see Section 8.3.

If a protocol amendment requires a change to a centre's Informed Consent Form, AstraZeneca/BIG/Partners, NRG Oncology/CTEP for US centres, and the centre's Ethics Committee are to approve the revised Informed Consent Form before the revised form is used.

If required by local regulations, any administrative changes will be communicated to or approved by each Ethics Committee.

#### 8.6 Audits and inspections

Authorised representatives of AstraZeneca, a regulatory authority, or an Ethics Committee may perform audits or inspections at the centre, including source data verification. The purpose of an audit or inspection is to systematically and independently examine all study-related activities and documents, to determine whether these activities were conducted, and data were recorded, analysed, and accurately reported according to the protocol, Good Clinical Practice (GCP), guidelines of the International Conference on Harmonisation (ICH), and any applicable regulatory requirements. The investigator/ site staff should contact the site monitor immediately if contacted by a regulatory agency about an inspection at the centre.

#### 9. STUDY MANAGEMENT

# 9.1 Pre-study activities

Before the first patient is entered into the study by a site, a representative of AstraZeneca/BIG/Partners may visit the investigational study site to:

• Determine the adequacy of the facilities

- Determine availability of appropriate patients for the study
- Discuss with the investigator(s) (and other personnel involved with the study) their responsibilities with regard to protocol adherence, and the responsibilities of AstraZeneca/BIG/Partners or representatives. This will be documented in a Clinical Study Agreement or equivalent.

# 9.2 Training of study site personnel

Before the first patient is entered into the study, AstraZeneca/BIG/Partners will review and discuss the requirements of the Clinical Study Protocol and related documents with the investigational staff and also train them in any study specific procedures and the WBDC.

The Principal Investigator should ensure that appropriate training relevant to the study is given to all site staff, and that any new information relevant to the performance of this study is forwarded to the staff involved.

The Principal Investigator will maintain a record of all individuals involved in the study (medical, nursing and other staff).

# 9.3 Monitoring of the study

During the study, a representative of AstraZeneca/BIG/Partners will have regular contacts with the study site, including visits to:

- Provide information and support to the investigator(s)
- Confirm that facilities remain acceptable
- Confirm that the investigational team is adhering to the protocol, that data are being accurately recorded in the eCRFs in a timely way, that biological samples are handled in accordance with the Laboratory Manual and that study drug accountability checks are being performed
- Perform source data verification (a comparison of the data in the eCRFs with the patient's medical records at the hospital or practice, and other records relevant to the study) including verification that the appropriate version of the consent form was used and that it was signed and dated prior to any study procedures. This will require direct access to all original records for each patient (e.g. clinic charts)
- If relevant, ensure withdrawal of informed consent to the use of the patient's biological samples is reported and biological samples are identified and disposed of/destroyed accordingly, and the action is documented, and reported to the patient.

The AstraZeneca/BIG/Partners representative will be available between visits if the investigator(s) or other staff at the centre needs information and advice about the study conduct.

#### 9.3.1 Source data

Refer to the Clinical Study Agreement or equivalent for location of source data.

# 9.4 Study agreements

The Principal Investigator at each centre should comply with all the terms, conditions, and obligations of the Clinical Study Agreement, or equivalent, for this study. In the event of any inconsistency between this Clinical Study Protocol and the Clinical Study Agreement, or equivalent, the terms of Clinical Study Protocol shall prevail with respect to the conduct of the study and the treatment of patients and in all other respects, not relating to study conduct or treatment of patients, the terms of the Clinical Study Agreement, or equivalent, shall prevail.

Agreements between AstraZeneca/BIG/NRG Oncology/Partners and the Principal Investigator should be in place before any study-related procedures can take place, or patients are enrolled.

#### 9.4.1 Archiving of study documents

The Investigator should follow the principles outlined in the Clinical Study Agreement (CSA) or equivalent.

# 9.5 Study timetable and end of study

The end of the study is defined as 'the last visit of the last patient undergoing the study'.

The study is expected to start in Q1 2014 and to end by 2028.

The study will end approximately 10 years following the randomisation of the last patient. Patients will be followed up until 10 years after the randomisation of the last patient.

The study may be prematurely terminated at individual centres if the study procedures are not being performed according to GCP, or if recruitment is slow. AstraZeneca may also terminate the entire study prematurely upon recommendations of the study IDMC if concerns for safety arise within this study or in any other study with olaparib.

# 10. DATA MANAGEMENT

Data management will be performed by Frontier Science.

The data collected through third party sources will be obtained and reconciled against study data by Frontier Science.

Adverse events and medical/surgical history will be classified according to the terminology of the latest version of the Medical Dictionary for Regulatory Activities (MedDRA).

Medications will be classified according to the AstraZeneca Drug Dictionary. Coding will be done by Frontier Science.

Additional details of data management procedures can be found in the Data Management Plan for the Study. This document will be continuously updated through the life of the study.

Data queries will be raised for inconsistent, impossible or missing data. All entries to the study database will be available in an audit trail.

The data will be validated as defined in the Data Management Plan. Quality control procedures will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. The Data Management Plan will also document the roles and responsibilities of the various functions and personnel involved in the data management process.

When all data have been coded, validated, and locked, clean file will be declared. Any treatment revealing data may thereafter be added and the final database will be locked.

The results from genetic research may be reported in the CSR for the main study, or in a separate report as appropriate. Refer to Appendix C.

# 11. EVALUATION AND CALCULATION OF VARIABLES

# 11.1 Calculation or derivation of efficacy variable(s)

# 11.1.1 Primary endpoint

The primary endpoint of the trial is invasive disease free survival (IDFS), defined as the time from randomisation to date of first recurrence, where recurrence is defined as loco-regional, distant recurrence, new cancer or death from any cause. IDFS is further detailed according to the standardised STEEP system definition (Hudis et al 2007) as one of the following:

- Ipsilateral invasive breast tumour recurrence (IIBTR): Invasive breast cancer involving the same breast parenchyma as the original primary.
- Regional invasive breast cancer recurrence: Invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast.
- Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or radiologically diagnosed as recurrent invasive breast cancer.
- Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
- Contralateral invasive breast cancer

 Second primary non-breast invasive malignancies (i.e., excluding new in situ carcinomas of any site). Second primary non-breast invasive malignancies include hematologic malignancies and MDS. Squamous or basal cell skin cancers will not be counted as primary endpoint events.

Loco-regional recurrence of the disease (ipsilateral or regional invasive breast cancer) should be cytologically/histologically confirmed. Appropriate imaging (CT, MRI bone and/or PET scan) of the chest/abdomen/pelvis or any other area as clinically indicated should be performed at the time of local recurrence to exclude further spread of the disease. Distant recurrence should be diagnosed by radiological examination and/or histopathological confirmation when metastatic lesion is easily accessible for biopsy.

For confirmed local recurrence events, the earliest date of diagnosis based on an objective finding (physical exam, radiological/imaging assessment, cytological/histopathological assessment) will be used to determine the time to event for the analysis but not the date of the first symptoms or blood analysis abnormality. For example if a physical exam results in 'suspected' disease recurrence and disease recurrence is then confirmed by cytology/histology then the date of the physical exam will be used to derive the time to event.

For confirmed distant recurrence the date of the earliest radiological/imaging examination or cytological/histopathological assessment linked to the diagnosis will be used to determine the time to event for the analysis (i.e. physical exam will not be considered within the derivation of time to distant recurrence nor will be symptoms or blood analysis).

Invasive contralateral breast cancer or invasive non-breast secondary primary cancer should be confirmed by histopathological report. The date of the earliest objective finding related to diagnosis of the new cancer will be used as the date of new cancer for the analysis.

If two recurrence events (local and distant) are reported within 2 months of each other then this is referred to as a simultaneous event and will be considered as a single event. In this situation the worst case will be taken as the event 'type' but the date of recurrence will be the earliest date of the two events. For example if local and distant recurrence are reported within a 2 month period then for the analysis and reporting of IDFS the event type will be distant recurrence but the date of recurrence will be the earliest date of the two events.

If two recurrence events are reported but more than 2 months has elapsed between the events then the events will be regarded as two separate recurrence events and the earliest event and corresponding date of event will be used in the derivation of IDFS (i.e. IDFS is based on the first recurrence event).

If a patient dies during the study with no documented disease recurrence or invasive contralateral breast cancer or invasive non-breast secondary primary cancer then death will be regarded as an event and the date of death will be used to determine the patients IDFS time.

Patients who have not had a recorded IDFS event at the time of the analysis will be censored at the date of their last disease evaluation. Disease evaluation includes mammogram and/or breast MRI (MRI preferred for patients younger than 50 years), other radiological/imaging examination or clinical examination (e.g. physical exam).

#### 11.1.2 Secondary endpoints

#### 11.1.2.1 Overall Survival

Overall survival is defined as the time from the date of randomisation until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.

#### 11.1.2.2 Distant disease free survival (DDFS)

DDFS will be defined as the time from randomisation until documented evidence of first distant recurrence of breast cancer. Distant recurrence will include the following events:

- Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or radiologically diagnosed as recurrent invasive breast cancer.
- Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
- Second primary non-breast invasive cancer.

Evidence of distant recurrence should be provided by either radiological examination or preferably by histopathological examination when metastasis is easily accessible for biopsy.

Second primary non-breast invasive cancer should be confirmed by histopathological report.

For the analysis of DDFS, the date of the confirmed DDFS event will use the earliest assessment date from the radiological and/or histological or cytological assessment. For example if a patient has distant recurrence suspected by radiological examination which is later confirmed by biopsy then the date of the radiological examination will be used as the date of event.

Patients who do not have documented evidence of DDFS at the time of the analysis of DDFS will be censored at the date of their last clinical examination (i.e. last physical exam or radiological evaluation).

The first site of distant recurrence will be recorded and used in the analysis. Information on subsequent sites of recurrence will also be collected during follow-up assessments to ensure as complete as possible information on distant recurrence is obtained.

# 11.1.2.3 Incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer

The incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer will each be considered separately and be defined as the number and percentage of patients with documented evidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer regardless of when this occurs (i.e. does not need to be their first recurrence event).

All patients should be followed for evidence of new primary breast cancers and all other cancers. This includes patients with a first event of local or distant recurrence as they may go on to develop new cancers in the future. All new cancers will be collected for all patients not just the first new cancer.

Data analyses of new contralateral breast cancer (invasive and non-invasive) will exclude patients who have had bilateral mastectomy prior to randomisation.

Data analyses of new ovarian cancers will exclude patients who have had both ovaries removed prior to randomisation.

Data analyses of new fallopian tube cancers will exclude patients who have had both fallopian tubes removed prior to randomisation.

Data analyses of new peritoneal cancer will include all patients in the ITT populations.

#### 11.2 Calculation or derivation of safety variable(s)

Safety and tolerability will be assessed in terms of AEs, deaths, laboratory data and vital signs. These will be collected for all patients. Appropriate summaries of these data will be presented as described in Section 12.

# 11.2.1 Other significant adverse events (OAE)

During the evaluation of the AE data, an AstraZeneca medically qualified expert will review the list of AEs that were not reported as SAEs and DAEs. Based on the expert's judgement, significant adverse events of particular clinical importance may, after consultation with the Global Patient Safety Physician, be considered OAEs and reported as such in the Clinical Study Report. A similar review of laboratory/vital signs/ECG data will be performed for identification of OAEs.

Examples of these are marked haematological and other laboratory abnormalities, and certain events that lead to intervention (other than those already classified as serious), dose reduction or significant additional treatment.

# 11.3 Calculation or derivation of patient reported outcome variables

Patient reported outcomes will be assessed based on the FACIT-Fatigue symptoms and the EORTC QLQ-C30 questionnaires. Further details are given in Section 12.2.3 and full details will be provided in the statistical analysis plan.

# 11.4 Calculation or derivation of pharmacokinetic variables

The pharmacokinetic (PK) analysis of the plasma concentration data for olaparib will be performed at AstraZeneca R&D or by a CRO identified by AstraZeneca R&D. The actual sampling times will be used in the PK calculations. For each patient providing a complete set of PK samples, non-linear mixed effects modelling (NONMEM) will be used to estimate steady state  $C_{max}$ , AUC and  $C_{min}$ .

# 11.5 Calculation or derivation of pharmacodynamic variable(s) - not applicable

# 11.6 Calculation or derivation of variables

Any data summaries that will be reported in the main clinical study report will be detailed within the statistical analysis plan. Additional exploratory analyses or data summaries that may be produced outside of the main study report will be defined in an exploratory analysis plan, if appropriate.

- 11.7 Calculation or derivation of health economic variables –not applicable
- 12. STATISTICAL METHODS AND SAMPLE SIZE DETERMINATION

# 12.1 Description of analysis sets

A comprehensive statistical analysis plan (SAP) will be prepared before first subject in (FSI).

Table 13 gives a summary of outcome variables and analysis populations.

#### 12.1.1 Full analysis set

Intention to treat (ITT): The primary statistical analysis of the efficacy of olaparib will include all randomised patients and will compare the treatment groups on the basis of randomised treatment, regardless of the treatment actually received. Patients who were randomised but did not subsequently go on to receive study treatment are included in the Full Analysis Set (FAS).

For the interim analysis two efficacy populations will be defined

1. ITT population: This will include all randomised patients and will compare the treatment groups on the basis of randomised treatment, regardless of the treatment actually received. Note: it is anticipated that all patients will be randomised by the time of the interim analysis.

2. Mature cohort ITT population: This will include the first 900 randomised patients only and will compare the treatment groups on the basis of randomised treatment, regardless of the treatment actually received.

#### 12.1.2 Safety analysis set

All patients who received at least one dose of randomised study treatment, olaparib or placebo, will be included in the safety analysis set. If a patient receives at least one dose of olaparib he/she will be summarised in the olaparib arm for safety summaries (e.g. olaparib arm will include patients randomised to olaparib who receive at least one dose of olaparib or placebo patients who receive at least one dose of olaparib in error at any time). If a patient randomised to olaparib receives only placebo treatment then he/she will be summarised as part of the placebo arm.

Table 13 Summary of Outcome Variables and Analysis Populations

| Outcome Variable | Populations |
|---|---|
| Efficacy Data - Interim | |
| IDFS | FAS (ITT), Mature cohort ITT |
| Other efficacy variables | FAS (ITT) |
| Efficacy data- Final | FAS (ITT) |
| IDFS, OS, DDFS, incidence of contralateral breast cancers, new primary ovarian, new primary fallopian tube cancers and new primary peritoneal cancer and symptom/HRQoL endpoints | |
| Demography | FAS (ITT) |
| Pharmacokinetics data | PK |
| Safety Data | |
| Exposure | Safety |
| Adverse Events | Safety |
| Lab measurements | Safety |
| Vital Signs | Safety |

#### 12.1.3 PK analysis set

PK data will be analysed according to treatment received. This population will comprise all randomised to olaparib patients who receive at least one dose of study treatment and have at least one PK sample collected.

# 12.2 Methods of statistical analysis

#### 12.2.1 Analysis of primary endpoint

# 12.2.1.1 Primary analysis

The primary analysis of IDFS will occur when a minimum of 330 IDFS events have been observed (to provide at least 90% power to detect a hazard ratio of 0.7). Based on the event rate from the 10 November 2017 database, the number of IDFS events required to trigger the primary analysis is expected to be accrued by November 2020 (80% CI: March 2020 to September 2021). The maturity rate will be 18.3%, where maturity is defined as the number of events divided by the total number of randomised patients.

IDFS will be compared across two treatment arms using a log rank test stratified by the stratification factors at randomization, and the corresponding p-value will be reported as the primary analysis result. In addition, IDFS will be analysed using a stratified Cox proportional hazard model stratified by the stratification factors at randomisation and using the Efron approach for handling ties. The point estimate of the treatment effect, i.e., the hazard ratio of IDFS (olaparib vs. placebo) will be obtained by maximizing the Cox partial likelihood function, which is the product of the partial likelihood of each stratum. The 95% confidence interval will be estimated using the profile likelihood approach.

A Kaplan-Meier plot of IDFS will be presented by treatment group. Summaries of the number and percentage of patients experiencing an IDFS event, and the type of event (recurrence or death) will be provided for each treatment.

The estimated 3 year IDFS will be summarised (using estimates from the KM curve) and presented by treatment group.

#### 12.2.1.2 Sensitivity analysis

If applicable, an analysis will be performed for IDFS using the same model as described above but based on all randomised patients confirmed to have gBRCA mutations by the central test. This analysis is only required if the analysis population differs from the primary ITT population.

Any patients mis-stratified in the randomisation system (i.e. incorrect details are entered at the time of randomisation) will be included in the primary stratified log rank test and Cox proportional hazard model using the baseline data collected from the randomisation system (Registration and Randomisation System). If >5% of randomised patients are incorrectly stratified (i.e., randomization system data does not match baseline data), then a sensitivity analysis will be performed for IDFS based on the (correct) baseline data collected in the eCRF. If the results of ER and PgR status from the local and central labs differ in >5% of randomised patients, a sensitivity analyses will also be performed based on ER and/or PgR positive/HER2 negative and TNBC subsets as defined by the central laboratory testing.

The assumption of proportionality will be assessed. Proportionality will be tested firstly by producing plots of complementary log-log (event times) versus log (time) and, if these raise concerns, a time dependent covariate would be fitted to assess the extent to which this represents random variation. Note that in the presence of non-proportionality, the HR will be interpreted as an average HR over the observed extent of follow-up.

As patients will be randomised, imbalances in demographic factors between the treatment groups are not anticipated. However if any imbalances should occur, these additional demographic variables may be fitted into the stratified Cox model. The HR and associated confidence interval would be presented.

#### 12.2.1.3 Subgroup analysis

Subgroup analyses will be conducted to assess consistency of treatment effect across potential or expected prognostic factors, including the baseline stratification factors.

If there are too few results available for a meaningful analysis of a particular subgroup (it is not considered appropriate to present analyses where there are less than 5 events in either treatment group), the relationship between that subgroup and IDFS will not be formally analysed. In this case, only descriptive summaries will be provided.

The following subgroups are of primary interest:

- Hormone receptor status (ER and/or PgR positive and HER2 negative; TNBC)
- Neoadjuvant chemotherapy; adjuvant chemotherapy
- Prior platinum therapy for current breast cancer (Yes;No)
- BRCA mutation type (BRCA1; BRCA2; BRCA1/2 both)
- Hormone receptor status by prior chemotherapy setting (if there are sufficient events to split into the four groups)
  - ER and/or PgR positive with neoadjuvant chemotherapy
  - ER and/or PgR positive with adjuvant chemotherapy
  - ER and PgR negative with neoadjuvant chemotherapy
  - ER and PgR negative with adjuvant chemotherapy
- BRCA status by prior platinum therapy setting
  - BRCA1 with prior platinum therapy for current breast cancer

- BRCA1 with no prior platinum therapy for current breast cancer
- BRCA2 with prior platinum therapy for current breast cancer
- BRCA2 with no prior platinum therapy for current breast cancer

The following additional subgroups will also be analysed to assess consistency in treatment effect across a broader set of baseline characteristics known before start of study medication:

- Type of prior Neo/Adjuvant chemotherapy (anthracycline; taxane; anthracycline plus taxane)
- Type of breast surgery prior to randomisation (breast conservation; unilateral mastectomy; bilateral mastectomy)
- Bilateral Oophorectomy (Yes; No)
- Axillary nodal status at surgery prior to randomisation (Positive or negative for the post adjuvant patients only)
- CPS+EG score at baseline (2, 3 or 4; 5 or 6 for the post neoadjuvant group only)
- Age at randomisation (<50; 50-64;  $\ge65$ )
- Race
- Sponsor (AZ; NRG Oncology)

Other baseline variables may also be assessed if there is clinical justification. These would be pre-defined within the SAP.

For each subgroup, the HRs (olaparib: placebo) and associated CIs will be calculated from a Cox proportional hazards model (using the Efron approach for handling ties) that contains the treatment term, factor and treatment-by-factor interaction term. The treatment effect HRs for each treatment comparison along with their confidence intervals will be obtained for each level of the subgroup from this single model. The HRs and 95% CIs will be presented on a forest plot including the HR and 95% CI from the overall population (using the primary analysis).

No adjustment to the significance level for testing subgroups will be made since all these subgroup analyses will be considered exploratory. The results would be used as supportive data for the primary analysis of IDFS based on all randomised patients.

# 12.2.1.4 Analysis of Interaction

The presence of quantitative interactions will be assessed by means of an overall global interaction test. This will be performed in the overall population by comparing the fit of a Cox proportional hazards model including treatment, all covariates (including stratification factors), and all covariate-by-treatment interaction terms, with one that excludes the interaction terms and will be assessed at the 2-sided 10% significance level. If a covariate does not have more than 20 events per level (of the covariate) it will be included as a covariate in the model, but the covariate-by-treatment interaction term will be omitted. If the fit of the model is not significantly improved then it will be concluded that overall the treatment effect is consistent across the subgroups.

If the global interaction test is found to be statistically significant, an attempt to determine the cause and type of interaction will be made. Stepwise backwards selection will be performed on the saturated model, whereby (using a 10% level throughout) the least significant interaction terms are removed one-by-one and any newly significant interactions re-included until a final model is reached where all included interactions are significant and all excluded interactions are non-significant. Throughout this process all main effects will be included in the model regardless of whether the corresponding interaction term is still present. This approach will identify the factors that independently alter the treatment effect and prevent identification of multiple correlated interactions.

Any quantitative interactions identified using this procedure will then be tested to rule out any qualitative interaction using the approach of Gail and Simon 1985.

#### 12.2.2 Analysis of secondary endpoints

#### **OS and DDFS**

OS and DDFS will be analysed at the time of the IDFS analysis as per the multiple testing procedure (MTP) outlined in Section 12.2.5 and will use the same methodology and model as described above for the primary analysis of IDFS.

If applicable, a sensitivity analysis will be performed for DDFS and OS using the same model as described above for IDFS but based on all randomised patients confirmed to have gBRCA mutations by the central test. This analysis is only required if the analysis population differs from the primary ITT population. Subgroup analyses will also be conducted for DDFS and OS based on the same subgroups described above for IDFS.

DDFS and OS will be analysed at the time of the primary analysis for IDFS (when 330 IDFS events are reported).

The final OS analysis will be conducted once the trial follow-up is complete (i.e. 10 years from when the last patient is randomised, estimated 14 years from first patient randomised assuming recruitment of 5 years).

In addition another analysis will be performed half way between the primary IDFS analysis and the final overall survival analysis (estimated around 10 years from first patient randomised but timings will be driven by the primary IDFS analysis once known). At this time point both DDFS and OS will be analysed and some alpha will be reserved for formal hypothesis testing. IDFS may also be updated if more information is available but this would be considered a supportive update of the primary analysis and no alpha will be reserved for IDFS

For details on alpha spend and how this will be allocated across the planned analyses see Section 12.2.6.

# Incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer

The actual number and percentage of patients with new contralateral breast cancers (invasive and non-invasive), new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancers will be presented. In addition a table summarising all reported new cancers (i.e. not just breast, ovarian, fallopian tube or peritoneal cancers) will also be produced.

As described in Section 11.1.2.3, patients who have had a bilateral mastectomy prior to randomisation will be excluded from the analysis of new contralateral breast cancers (invasive and non-invasive) and patients who have had a bilateral oophorectomy prior to randomisation will be excluded from the analysis of new ovarian cancers and patients who have had their fallopian tubes removed prior to randomisation will be excluded from the analysis of new fallopian tube cancers.

The cumulative incidence of new primary contralateral invasive breast, new primary contralateral non-invasive breast, new primary ovarian cancers, new primary fallopian tube cancers and new primary peritoneal cancers will be compared between treatment groups using competing risk analysis (Gray test, Fine and Gray 1999). Death will be considered a competing risk for each endpoint. In addition, bilateral mastectomy after randomization will be a competing risk for the contralateral breast cancer analyses, bilateral oophorectomy will be a competing risk for the new primary ovarian cancers analysis and removal of the fallopian tubes will be a competing risk for the new primary fallopian tube cancer analysis. Hazard ratios and 95% confidence intervals from competing risks regression analyses (Fine and Gray 1999) adjusted for treatment and the stratification factors will also be presented – more details of these analyses are given in the SAP (Edition 2).

#### Safety

Safety data will be summarised descriptively in terms of AEs, vital signs, clinical chemistry & haematology and physical exam and will include data from the treatment and safety follow-up period. Cumulative incidence plots may also be presented for specific adverse events or

groups events of interest. Further information on the summary of safety data will be provided in the SAP.

#### 12.2.3 Analysis of patient reported outcomes

#### 12.2.3.1 Hypotheses and objectives

The hypotheses and measurement strategy focus on the fact that patients in the trial will be starting with significant decrements in HRQoL and high rates of symptoms at study entry (baseline) due to previous chemotherapy and local treatments (surgery with or without radiation therapy). All analyses of Patient Reported Outcomes will be conducted on ITT population as listed in Table 13. Therefore, the following hypotheses are proposed, based on the expected toxicities of olaparib.

#### **Primary hypothesis**

Patients receiving olaparib may experience greater fatigue severity during treatment than those receiving placebo as measured by the FACIT-Fatigue scale at 6 and 12 months after randomisation

#### Secondary hypotheses

Patients receiving olaparib may experience greater GI symptoms (nausea, vomiting and diarrhoea) severity during treatment than those receiving placebo as measured at 6 and 12 months after randomisation but no difference expected by 24 months after randomisation.

There will be no difference in fatigue post discontinuation of study treatment as measured at 18 and 24 months.

There will be no difference in QOL between the two treatment arms as measured by the global QOL score and other sub scales from the EORTC QLQ-C30 at 6, 12, 18 and 24 months after randomisation and patients will demonstrate improvements in functioning over time.

#### **Primary PRO objective**

To determine the effect of olaparib on patient-reported fatigue at 6 and 12 months after randomisation as measured by the FACIT-Fatigue symptoms questionnaire.

#### **Secondary PRO objectives**

- To determine the effect of olaparib on patient-reported GI symptoms (nausea, vomiting and diarrhea) over time at 6, 12, 18 and 24 months as measured by the EORTC QLQ-C30 scale.
- To determine the effect of olaparib on patient reported fatigue over time at 6, 12, 18 and 24 months as measured by the FACIT-Fatigue questionnaire.

- To determine if there will be a difference in QOL between the two treatment groups over time as measured by the 2 item global QOL score of the EORTC QLQ-C30 scale at 6, 12, 18 and 24 months and assess if patients demonstrate improvement in scores over time.
- To examine and compare the effect of olaparib over time on different functional sub scale scores as measured by the EORTC QLQ-C30 and assess if patients demonstrate improvement in functioning over time, with particular interest in the physical and emotional sub scales.

#### 12.2.3.2 Statistical considerations for patient reported outcomes

# Statistical analyses

# Primary endpoint - Fatigue

For the primary hypothesis, the composite fatigue score (FACIT-Fatigue questionnaire) measured at 6 and 12 months after randomisation will be compared between the two treatment arms using analysis of covariance (ANCOVA) with adjustment for the corresponding baseline measurement. Separate analyses will be done for patients who have received prior neoadjuvant chemotherapy and patients who have received standard post-surgical adjuvant chemotherapy. Separate analyses are preferable because the timing of chemotherapy is expected to impact the fatigue outcome directly. Each comparison will be performed at the significance level of 0.05. No multiple comparisons adjustment will be employed since these outcomes evaluate the toxicity of the study treatment.

To further assess the effect of olaparib on fatigue over time (study treatment period and the year following) the composite fatigue score (FACIT-Fatigue questionnaire) measured at 6, 12, 18 and 24 months after randomisation will be compared between the two treatment arms using a mixed model for repeated measures (MMRM) analysis of all of the post baseline scores. The model will include treatment, time and treatment by time interaction as explanatory variables and baseline score and baseline by time interaction as covariates. The treatment by visit interaction will remain in the model regardless of significance. The adjusted mean change from baseline estimates for each treatment arm, difference in the adjusted mean change from baseline estimates between the arms and corresponding confidence intervals will be presented by time point. Plots of the adjusted means changes over time will also be presented.

# **Secondary PRO endpoints**

A secondary analysis based on GI symptoms (nausea, vomiting and diarrhoea) over time from the EORTC QLQ-C30 scale will be performed using the same MMRM model described above. The adjusted mean change from baseline estimates for each treatment arm, difference in the adjusted mean change from baseline estimates between the arms and corresponding confidence intervals will be presented by visit. Plots of the adjusted means changes over time will also be presented for nausea, vomiting and diarrhoea.

To assess if there are any difference in HRQoL, the 2 item global QOL score assessed by EORTC QLQ-30 measured at 6, 12, 18 and 24 months after randomisation will be compared between the two treatment arms using the same MMRM model described above. Plots over time will also be produced for the global QOL score.

In addition, other subscales of the EORTC QLQ-C30 will be analysed using the MMRM model described above with particular interest in the emotional and physical subscales. Plots over time will also be produced.

All secondary analyses are considered exploratory and therefore no adjustments for multiplicity will be made. For each comparison, p-values (along with CIs) will be generated to help aid interpretation of the results using a nominal significance level of 0.05 (2-sided).

Because this trial is being conducted internationally, responses to patient reported outcomes may be influenced by differences between country/language categories (Bernhard J et al 2007). Therefore, analyses will be stratified by country/language groups. Further details will be provided in the SAP.

Adjustment for previous treatment exposures (radiation, type of chemotherapy, and surgery) may also be considered as part of the secondary analyses. Further details will be given in the SAP

#### Sample size consideration

We assume that half of triple negative patients and a quarter of hormone receptor positive patients will have received neoadjuvant chemotherapy and we anticipate that 95% of patients enrolled in the trial will complete the HRQoL instrument. In addition, adjusting downward to allow for 20% of missing data at the 12 months assessment point, we expect that data from 633 neoadjuvant and 735 adjuvant patients will be available (assuming that 15% of the total 1800 enrolled patients are ER and/or PgR positive HER2 negative). These will be sufficient to provide statistical power of 93% and 96% correspondingly to detect a difference of 3 points on the FACIT-Fatigue scale score between treatment groups assuming a standard deviation of 10.9 (Cella D et al 2002) (estimated SD of mean baseline score) and controlling  $\alpha$ -level at 0.05. A collection of PROs and QOL from all patients enrolled in the main trial will give us sufficient statistical power to detect important differences between two treatment groups.

#### Missing PRO data

A certain amount of missing data is expected. If data for individual items are missing, imputation will be done as follows: if less than 50% of the subscale items were missing (e.g. at most 2 out of 5 items, etc), the subscale score based on the non-missing items will be divided by the number of non-missing items and multiplied by the total number of items on the subscale. If at least 50% of the items are missing, that subscale will be treated as missing (not evaluable). If the scale is a single-item measure, a missing value will automatically be defined as 'Non-Evaluable'. The information from patients with missing data will be reviewed

in order to determine whether data analytic procedures are likely to be biased. Patients with missing data will be reviewed for imbalances in factors such as trial arm, treatment adherence, institution, and reason for non-adherence. When QOL data are missing at a particular time point, data from prior time points will be reviewed in order to investigate whether missing status was preceded by a significant change in QOL scores. In addition, we will investigate whether missing item status is related to other scores on the same questionnaire. If no missing data mechanism can be detected following this review, the data will be analysed assuming the data are missing at random. If, on the other hand, a missing data mechanism appears to be present, we will undertake to develop an appropriate analytic strategy to control for the potential bias and, if possible, to impute the missing values. We will also present sensitivity analyses based on varying assumptions about the missing-data mechanism.

Full details on the analysis and derivation of PRO endpoints will be provided in the statistical analysis plan (SAP).

#### 12.2.3.3 Pharmacokinetic analysis

The plasma concentration-time data will be analysed by non-linear mixed effects modelling in order to evaluate the pharmacokinetic characteristics of olaparib, quantify variability in the pharmacokinetics, identify demographic or pathophysiological covariates which may explain the observed variability and explore exposure-response relationships.

The olaparib plasma concentration data obtained from the samples collected in this study will be included in the listings of the CSR but these data will be pooled with data from other studies in order to perform a population PK analysis. The results of this analysis will be reported in a separate population PK report.





#### 12.2.5 Multiplicity strategy for primary and key secondary endpoints

The primary endpoint of the study is IDFS. However, key secondary endpoints will be OS and DDFS.

In order to describe the nature of the benefits of olaparib treatment IDFS, DDFS and OS will be tested at a 2-sided significance level of 5%.

However, in addition, in order to strongly control the overall type I error at 2.5% 1-sided, a multiple testing procedure (MTP) will be employed across the primary endpoint and all key secondary endpoints intended for label claims (DDFS and OS). The MTP will account for any interim analyses on IDFS, DDFS and OS and also planned further analyses post the primary IDFS analysis data cut off.

A hierarchical testing strategy will be employed where IDFS is tested first using the full test mass (i.e. full 2.5%, 1-sided alpha), then DDFS and OS will be tested if IDFS is significant based on a weighted proportion of the test mass (2% for DDFS and 0.5% for OS, 1-sided) which can be recycled to secondary endpoints not yet rejected. Testing stops when the entire test mass is allocated to non-rejected endpoints.

Figure 3 Multiple testing procedure



IDFS is planned to be analysed at the interim and the final analysis (see Section 12.2.6 for further details). If IDFS is significant at the interim based on the ITT population then secondary endpoints will be formally tested at the interim based on the MTP outlined above. To account for multiple analyses on each endpoint a separate alpha spending function will be applied to each endpoint (Glimm et al 2010). Further analyses of DDFS and OS with more mature follow-up may be required for which some alpha will be reserved for significance testing.

# 12.2.6 Interim analysis

A superiority interim analysis of IDFS will occur when half the events needed for at least 90% power (165 events) have been observed from the first 50% of patients recruited (i.e. from first 900 patients) providing a cohort of patients with a similar level of maturity that is planned for the final analysis. Based on the database at time of amendment, the interim analysis is predicted to be October 2019 (80% CI: March 2019 to August 2020). The predictions will be tracked and monitored as more patients are enrolled in the study and additional data is added to the database. Two populations will be analysed at the interim analysis based on the analysis methods described in Section 12.2.1 for IDFS

- Primary: ITT population (all patients randomised, estimated 254 events [80% CI: 226 to 289])
- 2 Supportive: Mature cohort population (first 900 patients randomised, 165 events anticipated)

The inclusion of a mature cohort population at the interim is to provide confidence that any observed treatment effect from the interim ITT population is maintained with longer-term

follow-up. It is anticipated, based on the assumed recruitment and event rate that the interim analysis will occur approximately 5.3 years after the first patient is randomised and that all patients will have been randomised. At the time of the interim analysis, median time at risk per patient is expected to be 27 months in the ITT set, and 34 months in the mature cohort. The critical HR value at the interim analysis is 0.701.

Evidence of superiority for IDFS would only be determined at the interim if the results from both analysis populations provide evidence of a sustainable clinically relevant treatment effect for IDFS. More specifically, as a minimum the result in the ITT population would need to have met the statistical threshold defined below. Having met the statistical threshold in the ITT population, the result in the mature cohort (i.e. HR) would need to be of a similar magnitude such that the IDMC would consider it supportive of the ITT result and therefore have added confidence in the result in the ITT population. Statistical significance is not required for the mature cohort population. This analysis will be regarded as supportive, based on a cohort of patients with longer-term follow-up, to aid interpretation of the result in the ITT population based on interim data. Other outcome measures such as 3 year IDFS rate will also be presented to aid the interpretation of the HRs (particularly in the case where the assumption of proportional hazards may not hold). KM plots will also be produced for IDFS.

The test mass alpha for IDFS (1 sided 2.5%) will be split between the final and the interim analysis using a bespoke spending function where a fixed significance level will be assigned at the interim and the remaining significance level assigned to the final analysis, taking account of correlation (Stone 2010). A 2-sided significance level of 0.005 will be assigned to the interim analysis so that a highly significant and clinically relevant result will need to be observed to declare superiority on IDFS. As an illustration, if 70% of the total required 330 IDFS events have occurred in the ITT population at the interim then the observed HR would need to be <0.7 for superiority to be declared. The HR in the mature cohort would need to be supportive of the ITT result. More detail around the criteria required for the mature cohort will be provided in the IDMC charter or SAP.

If the null hypothesis for IDFS is rejected at the interim for the ITT population then secondary endpoints (DDFS and OS) will be tested based on the MTP procedure outlined in Section 12.2.5 using the significance levels provided in Table 14. If IDFS is not significant at the interim, DDFS and OS will not be tested at the IDFS interim and the significance level allocated to the IDFS interim for DDFS and OS will not be allocated to later timepoints.

Similar to IDFS, a bespoke spending function will be applied to the secondary endpoints OS and DDFS where a fixed significance level will be assigned to each analysis time point and the remaining significance level assigned to the final analysis time point controlling the overall type 1 error at the pre-specified alpha amount (Stone 2010). Provided the last analysis is known in advance of the penultimate one then the remaining alpha can be split to ensure that some alpha is always reserved for the final analysis. This approach allows flexibility in the number of analyses while appropriately controlling the overall type 1 error. Three analyses are planned for DDFS and four for OS for which some alpha will be reserved for significance

testing. If additional analyses are required beyond the planned analyses and some alpha is still available for testing then any remaining alpha can be further split to strongly control the type 1 error (based on process described above). If no alpha remains then the additional analyses will be considered supportive updates of the already conducted analyses.

Given the split in alpha between DDFS and OS, if OS is significant based on the assigned significance level then the alpha assigned to OS will be recycled to DDFS and split across the planned analyses (and vice versa if DDFS is significant alpha for DDFS will be recycled to OS and split across analyses). The recycled alpha will be split based on the ratio of the originally assigned alpha split. For example if the original alpha allocation was split 1/3 for each analysis time point then the recycled alpha would also be split 1/3 across each analysis time point. For example, at the first interim analysis, assume IDFS is statistically significant and the secondary endpoint OS is also statistically significant. The significance level for testing DDFS is therefore  $0.005 + (\text{alpha assigned to OS recycled to DDFS and split across the planned analyses), i.e. <math>0.005 + (1\% * 0.005/0.04 = 0.00125) = 0.00625$ , or alternatively thought of as 0.005 \* 5/4.

Secondary endpoints will be assessed based on the ITT population. Table 14 shows the different 2-sided significance levels that will be applied to the primary and secondary endpoints across the planned analyses as well as the total alpha spend for each endpoint. Note the significance level for the final analyses of each endpoint will be calculated using the relevant correlation based on the actual number of events for each analysis, the previous alpha spend and the total allocated alpha for that endpoint.

Table 14 Summary of 2-sided significance levels and total alpha spend across the endpoints and analyses

| Endpoints | Interim<br>analysis | Final IDFS<br>analysis | DDFS and OS analysis | Final OS<br>analysis | |
|---|---|---|---|---|---|
| Estimated timings from FSI** | 5.3 years | 6.5 years | 10 years | 14 years | |
| | Significance level | Significance level | Significance level | Significance level | Total<br>alpha<br>spend (2-<br>sided) |
| IDFS | 0.005 | TBC* | N/A | N/A | 5% |
| If IDFS is state analysis | istically significan | t and alpha is not recyc | cled between second | dary endpoints | at the |
| DDFS | 0.005 | 0.02 | TBC* | N/A | 4% |
| OS | 0.002 | 0.003 | 0.004 | TBC* | 1% |

If IDFS is statistically significant and alpha is recycled between secondary endpoints at the analysis

Date 18 May 2018

Table 14 Summary of 2-sided significance levels and total alpha spend across the endpoints and analyses

| Endpoints | Interim<br>analysis | Final IDFS<br>analysis | DDFS and OS analysis | Final OS<br>analysis | |
|---|---|---|---|---|---|
| Estimated timings from FSI** | 5.3 years | 6.5 years | 10 years | 14 years | |
| DDFS | 0.00625 | 0.025 | TBC* | N/A | 5% |
| OS | 0.01 | 0.015 | 0.02 | TBC* | 5% |

<sup>\*</sup>TBC: to be calculated; significance level to be calculated once relevant correlation based on the actual number of events for each analysis is known taking account of previous alpha spend and total allocated alpha \*\*FSI: first subject in

The IDMC will review the data from the interim analysis. The boundaries defined by the interim p-values for efficacy will be used as guidelines by the IDMC along with all other relevant trial information, including the safety data, to decide if it is appropriate to make a recommendation other than that to continue the trial as planned.

At the time of the interim analysis for superiority, an assessment of futility will also be performed. This futility assessment will be based on the probability of eventually showing statistical significance for the primary endpoint when the final number of IDFS events (n=330) is reached (Lachin 2005). The determination of this probability will be conditional on the observed data in the ITT population at the time of the interim analysis for superiority and on the assumed hazard ratio for the alternative hypothesis (IDFS HR=0.7). If the probability is less than 0.1, the IDMC will consider the option of declaring futility.

Full details on the process around the interim analysis and the efficacy criteria will be documented in the SAP and IDMC charter.

#### 12.2.7 Sample size justification

The primary endpoint of the study is IDFS and patients will be randomised 1:1 to either olaparib 300 mg b.i.d. (twice daily) or matching placebo.

A total of 1800 patients will be randomised into the study to achieve 330 IDFS events. If the true HR for the comparison of olaparib versus placebo in terms of IDFS is 0.7 then with 330 events, the analysis of IDFS will have 90% power to demonstrate a statistically significant difference in IDFS, assuming a 2-sided 5% significance level. The critical HR value at the primary analysis is 0.805.

The actual accrual pattern between June 2014 and February 2018 is shown in Table 15. It is estimated that 1800 patients will be randomised by April/May 2019 so that the study will take
approximately 5 years to complete recruitment (approximately 230 patients in US and approximately 1570 patients in the Rest of the World countries).

Table 15 Actual accrual between June 2014 and February 2018

| Interval since start of randomisation (months) | Number of patients randomised in interval | Cumulative number of patients randomised | Average number of patients randomised per month in interval |
|---|---|---|---|
| 0-6 | 21 | 21 | 3.5 |
| 6-12 | 94 | 115 | 15.7 |
| 12-18 | 174 | 289 | 29 |
| 18-24 | 180 | 469 | 33 |
| 24-30 | 229 | 698 | 38.2 |
| 30-36 | 249 | 947 | 41.5 |
| 36-42 | 234 | 1181 | 39 |
| 42-45* | 118 | 1299 | 39.3 |

\*Note: 3-month interval: December 2017 to February 2018 inclusive.

The primary analysis population will be all patients randomised (ITT). A subgroup analysis based on prior chemotherapy (adjuvant or neoadjuvant), prior platinum therapy (yes or no) and hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC) will be conducted to check for consistency in the treatment effect but this analysis is considered supportive of the primary analysis in the overall population.

During the trial, the Steering Committee will monitor the recruited patient population and actual event rate whilst remaining blinded to treatment. If the data suggests that the original sample size assumptions are incorrect such that achieving the required number of events with the current number of patients does not seem feasible then in consultation with the IDMC a decision may be made to increase the number of patients recruited into the trial to achieve the required 330 events.

## 12.3 Independent Data monitoring committee

This study will utilise an Independent Data Monitoring Committee (IDMC) whose members include therapeutic area experts and statisticians who are not employed by AstraZeneca and do not have any major conflict of interest. Members of the IDMC will be jointly selected by BIG, AstraZeneca, CTEP and NRG Oncology and the IDMC will report their recommendations to the Steering Committee.

The IDMC will meet approximately every 6 months and will review ongoing study progress including safety and, when appropriate, efficacy data. They will also review the data presented at the time of the protocol-defined interim analysis. The IDMC will have the ability to

recommend suspension of enrolment if safety concerns are identified at any of the 6 monthly assessments. At the interim analysis, both efficacy and safety will be reviewed and trial recommendations will be based on the totality of the data. The IDMC can recommend changes to the trial, including stopping of the trial, if they have concerns over the benefit risk profile for olaparib.

Reports for the IDMC will be prepared by an Independent Statistical Centre (ISC) and will be presented to the IDMC in closed session. Following review of data, the IDMC will make a recommendation regarding the future conduct of the trial to the Steering Committee. The IDMC recommendation will not contain any unblinded information or any information related to treatment outcomes of the trial.

A separate IDMC Charter will be developed defining the responsibilities and procedures for the IDMC.

# 13. IMPORTANT MEDICAL PROCEDURES TO BE FOLLOWED BY THE INVESTIGATOR

# 13.1 Medical emergencies and contacts

The Principal Investigator is responsible for ensuring that procedures and expertise are available to handle medical emergencies during the study. A medical emergency usually constitutes an SAE and is to be reported as such, see Section 6.4.4.

In the case of a medical emergency the investigator may contact Study Physician or Medical Team.

| Name | Role in the study | Address & telephone number |
|---|---|---|
| | Global Study Leader<br>responsible for the protocol at<br>central R&D site | AstraZeneca Pharma Poland |
| | Study Physician responsible<br>for the protocol at central<br>R&D site | AstraZeneca |
| | Global Safety Physician | AstraZeneca |
| Medical Team on behalf of the<br>Breast International Group<br>(BIG): | Responsible for handling on-study medical review, medical queries and participate in medical development of the protocol | BIG headquarters olympia.science@bordet.be |
| | Clinical Scientist<br>Medical Advisor<br>Medical Advisor | |

#### 13.2 Overdose

There is currently no specific treatment in the event of overdose with olaparib and possible symptoms of overdose are not established. Study treatment must only be used in accordance with the dosing recommendations in this protocol. Any dose or frequency of dosing that exceeds the dosing regimen specified in this protocol should be reported as an overdose. Monitors should report any overdose as a minor protocol deviation. The MTD is 300 mg b.i.d (tablet).

Adverse reactions associated with overdose should be treated symptomatically and should be managed appropriately.

- An overdose with associated AEs is recorded as the AE diagnosis/symptoms on the relevant AE modules in the eCRF and on the Overdose eCRF module.
- An overdose without associated symptoms is only reported on the Overdose eCRF module.

If an overdose on an AstraZeneca study drug occurs in the course of the study, then Investigators or other site personnel inform appropriate medical representatives immediately, or no later than 24 hours of when he or she becomes aware of it.

The designated study representative works with the Investigator to ensure that all relevant information is provided to the AstraZeneca Patient Safety data entry site.

For overdoses associated with SAE, standard reporting timelines apply (see Section 6.4.4). For other overdoses, reporting should be done within 30 days.

## 13.3 Pregnancy

All outcomes of pregnancy should be reported to AstraZeneca (see Table 16 and Table 17).

## 13.3.1 Maternal exposure

If a patient becomes pregnant during the course of the study the investigational product should be discontinued immediately.

The outcomes of any conception occurring from the date of the first dose of study medication until 3 months after the last dose of study medication must be followed up and documented.

Pregnancy itself is not regarded as an adverse event unless there is a suspicion that the investigational product under study may have interfered with the effectiveness of a contraceptive medication. Congenital abnormalities/birth defects and spontaneous miscarriages should be reported and handled as SAEs. Elective abortions without complications should not be handled as AEs. The outcome of all pregnancies (spontaneous

miscarriage, elective termination, ectopic pregnancy, normal birth or congenital abnormality) should be followed up and documented even if the patient was discontinued from the study.

If any pregnancy occurs in the course of the study, then Investigators or other site personnel inform appropriate medical representatives immediately, or no later than 24 hours of when he or she becomes aware of it.

The designated study representative works with the Investigator to ensure that all relevant information is provided to the AstraZeneca Patient Safety data entry site within 1 or 5 days for SAEs (see Section 6.4.4) and within 30 days for all other pregnancies.

The same timelines apply when outcome information is available.

The relevant module in the eCRF is used to report the pregnancy and the relevant eCRF module is used to report the outcome of the pregnancy.

## 13.3.2 Paternal exposure

Male patients should refrain from fathering a child or donating sperm during the study treatment period and for 3 months following the last dose. Pregnancy of the patient's partners is not considered to be an adverse event. However, the outcome of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal birth or congenital abnormality) should if possible be followed up and documented.

The outcome of any conception occurring from the date of the first dose until 3 months after the last dose should be followed up and documented.

Table 16 Pregnancy reporting and handling according to time of diagnosis

| Time point of diagnosis | Handling and reporting |
|---|---|
| During screening | Do not randomise, record as reason for screen failure by completing the Step 3 Screening Failure Confirmation checklist in the FS Registration and Randomisation system. |
| After randomisation but before first dose | Do not start study treatment, continue to follow patient for study end-points, report in eCRF and AstraZeneca Patient Safety DES via the paper Pregnancy form within 24 hours |
| During study treatment (maternal exposure) <sup>a</sup> | Discontinue from study treatment immediately, continue to follow patient for study end-points, report in eCRF, to medical team via email and AstraZeneca Patient Safety DES via the paper Pregnancy form within 24 hours |

Table 16 Pregnancy reporting and handling according to time of diagnosis

| Time point of diagnosis | Handling and reporting |
|---|---|
| Follow-up: Within 3 months of the end of study treatment | Continue to follow patient for study end-points, report in eCRF, to medical team via email and AstraZeneca Patient Safety DES via the paper Pregnancy form within 24 hours |
| Follow-up: After 3 months of the end of study treatment | Report in eCRF and to AstraZeneca Patient<br>Safety DES via the paper Pregnancy form within<br>30 days |

This includes pregnancies identified during Follow-up but with a probable date of conception during the period in which the patient was still receiving study treatment.

Table 17 Reporting outcomes of pregnancy according to time of diagnosis

| Time point of diagnosis | Normal outcome | Abnormal outcome <sup>a, b</sup> |
|---|---|---|
| During screening | No need to report on outcomes | No need to report on outcomes |
| After randomisation but before first dose | In eCRF and AstraZeneca Patient Safety<br>DES via the paper Pregnancy form Part II<br>within 30 days | Treat as an SAE (report within 24 hours) |
| During study treatment (maternal exposure) <sup>a</sup> | In eCRF, to the medical team via email<br>and AstraZeneca Patient Safety DES via<br>the paper Pregnancy form Part II within<br>24 hours | Treat as an SAE (report within 24 hours) |
| Follow-up: Within 3 months of the end of study treatment | In eCRF, to the medical team via email<br>and AstraZeneca Patient Safety DES via<br>the paper Pregnancy form Part II within<br>24 hours | Treat as an SAE (report within 24 hours) |
| Follow-up: After 3 months of the end of study treatment | In eCRF and AstraZeneca Patient Safety<br>DES via the paper Pregnancy form Part II<br>within 30 days | Treat as an SAE (report within 24 hours) |

Abnormal outcome means congenital abnormalities/birth defects, ectopic pregnancy and spontaneous miscarriages. Elective abortions without complications should not be handled as AEs.

If there is a suspicion that the investigational product under study may have interfered with the effectiveness of a contraceptive medication, pregnancy should be reported as an AE.

#### 14. LIST OF REFERENCES

#### Aaronson et al 1993

Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology.

#### Aebi et al 2011

S. Aebi, T. Davidson, G. Gruber & F. Cardoso. Primary breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Annals of Oncology 22 (Supplement 6): vi12–vi24, 2011.

## **American Cancer Society 2013**

American Cancer Society. Cancer Facts and Figures 2013. Atlanta, Georgia: American Cancer Society, 2013. http://www.cancer.org.

#### Antoniou et al 2003

Antoniou A, Pharoah PD, Narod S, Risch HA, Eyfjord JE, Hopper JL, et al. Average risks of breast and ovarian cancer associated with *BRCA*1 or *BRCA*2 mutations detected in case Series unselected for family history: a combined analysis of 22 studies. Am J Hum Genet 2003;72(5):1117-30.

#### Arun et al 2011

Arun B, Bayraktar S, Liu DD, Gutierrez Barrera AM, Atchley D, Pusztai L, et al. Response to neoadjuvant systemic therapy for breast cancer in *BRCA* mutation carriers and non-carriers: a single-institution experience. J Clin Oncol 2011; 29(28):3739-46.

#### Atchley et al 2008

Atchley DP, Albarracin CT, Lopez A, Valero V, Amos CI, Gonzalez-Angulo AM, et al. Clinical and pathologic characteristics of patients with *BRCA*-positive and *BRCA*-negative breast cancer. J Clin Oncol. 2008;26(26):4282-8.

## Bergfeldt et al 1995

Bergfeldt K, Einhorn S, Rosendahl I, Hall P. Increased risk of second primary malignancies in patients with gynecological cancer. A Swedish record-linkage study. Acta Oncol. 1995;34(6):771-7.

## Bernhard J et al 2007

Bernhard J, Zahrieh D, Castiglione-Gertsch M, et al. Adjuvant chemotherapy followed by goserelin compared with either modality alone: the impact on amenorrhea, hot flashes, and quality of life in premenopausal patients—the International Breast Cancer Study Group Trial VIII. J Clin Oncol 2007; 25:263-270.

#### Bordeleau et al 2011

Bordeleau L, Lipscombe L, Lubinski J, et al. Diabetes and breast cancer among women with *BRCA*1 and *BRCA*2 mutations. Cancer 2011;117:1812-8.

#### Bower et al 2000

Bower JE, Ganz PA, Desmond KA, et al. Fatigue in breast cancer survivors: occurrence, correlates, and impact on quality of life. J Clin Oncol 2000; 18(4):743-753.

#### Bower et al 2006

Bower JE, Ganz PA, Desmond KA, et al. Fatigue in long-term breast carcinoma survivors: a longitudinal investigation. Cancer 2006; 106(4):751-758.

#### Burnell et al 2010

Burnell M, Levine MN, Chapman JW, Bramwell V, Gelmon K, Walley B, et al. Cyclophosphamide, Epirubicin, and Fluorouracil Versus Dose-Dense Epirubicin and Cyclophosphamide Followed by Paclitaxel Versus Doxorubicin and Cyclophosphamide Followed by Paclitaxel in Node-Positive or High-Risk Node-Negative Breast Cancer. Journal of Clinical Oncology;vol28 no 1.

#### Cameron et al 2013

Cameron D, Brown J, Dent R et al. Adjuvant bevacizumab-containing therapy in triple-negative breast cancer (BEATRICE): primary results of a randomised, phase 3 trial. Lancet Oncol 2013; 14:933-42.

## **Carey 2011**

Carey LA. Directed Therapy of Subtypes of Triple-Negative Breast Cancer. The Oncologist 2011;16(suppl 1):71–78.

## Cella D et al 2002

Cella D, Eton DT, Lai JS, et al. Combining anchor and distribution-based methods to derive minimal clinically important differences on the Functional Assessment of Cancer Therapy (FACT) anemia and fatigue scales. J Pain Symptom Manage 2002; 24(6):547-561

## Cole and Strair 2010

Cole M, Strair R. Acute myelogenous leukemia and myelodysplasia secondary to breast cancer treatment: case studies and literature review. Am J Med Sci 2010;339(1):36-40.

#### Cortazar et al 2014

Cortazar P, Zhang L, Untch M, et al. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet 2014; 384:164-72.

#### Dent et al 2007

Dent R, Trudeau M, Pritchard KI, Hanna WM, Kahn HK, Sawka CA, Lickley LA, Rawlinson E, Sun P, Narod SA. Triple-negative breast cancer: clinical features and patterns of recurrence. Clin Cancer Res. 2007;13:4429-34.

## Fine and Gray 1999

Fine, J. and Gray, R. A Proportional Hazards Model for the Subdistribution of a Competing Risk, Journal of the American Statistical Association, 1999: 94, 496–509.

# Fong et al 2009

Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, et al. Inhibition of poly(ADP-ribose) polymerase in tumors from *BRCA* mutation carriers. N Engl J Med. 2009;361(2);123-34.

#### Foulkes et al 2010

Foulkes, W, Smith, IE, Reis-Filho, JS. Triple Negative Breast Cancer. N Engl J Med 2010;363;1938-48.

## Fowble et al 2001

Fowble B, Hanlon A, Freedman G, Nocolaou N, Anderson P. Second cancers after conservative surgery and radiation for stages I-II breast cancer: identifying a subset of women at increased risk. Int J Radiat Oncol, Biol, Phys. 2001; 51 (3);679-690.

## Gail and Simon 1985

Gail M, Simon R. Testing for qualitative interactions between treatment effects and patient subsets. Biometrics 1985;41:361-72.

#### Ganz et al 1998A

Ganz PA, Rowland JH, Desmond K, et al. Life after breast cancer: understanding women's health-related quality of life and sexual functioning. J Clin Oncol 1998; 16(2):501-514.

## Ganz et al 1998B

Ganz PA, Rowland JH, Meyerowitz BE, et al. Impact of different adjuvant therapy strategies on quality of life in breast cancer survivors. Recent Results Cancer Res 1998; 152(9):396-411.

#### Ganz et al 2002

Ganz PA, Desmond KA, Leedham B, et al. Quality of life in long-term, disease-free survivors of breast cancer: a follow-up study. J Natl Cancer Inst 2002; 94(1):39-49.

#### Ganz et al 2004

Ganz PA, Kwan L, Stanton AL, et al. Quality of life at the end of primary treatment of breast cancer: first results from the moving beyond cancer randomized trial. J Natl Cancer Inst 2004; 96(5):376-387.

#### Ganz et al 2011A

Ganz PA, Land SR, Geyer CE, et al. Menstrual history and quality-of-life outcomes in women with node-positive breast cancer treated with adjuvant therapy on the NSABP B-30 trial. J Clin Oncol 2011; 29(9):1110-1116.

#### Ganz et al 2011B

Ganz PA, Kwan L, Stanton AL, et al. Physical and psychosocial recovery in the year after primary treatment of breast cancer. J Clin Oncol 2011; 29(9):1101-1109.

## Gaymes et al 2008

Gaymes TJ, Shall S, MacPherson LJ, Twine NA, Lea NC, Farzaneh F, and Mufti GJ. Inhibitors of poly ADP-ribose polymerase (PARP) induce apoptosis of myeloid leukemic cells: potential for therapy of myeloid leukemia and myelodysplastic syndromes. Haematologica 2009; 94:638-646. doi:10.3324/haematol.2008.001933.

#### Gelmon et al 2011

Gelmon KA, Tischkowitz M, Mackay H, Swenerton K, Robidoux A, Tonkin K, et al. Olaparib in patients with recurrent high-grade serous or poorly differentiated ovarian carcinoma or triple-negative breast cancer: a phase 2, multicentre, open-label, non-randomised study. Lancet Oncol 2011; 12: 852–61

## Ginsburg et al 2010

Ginsburg OM, Kim-Sing C, Foulkes WD, Ghadirian P, Lynch HT, Sun P, et al. *BRCA*1 and *BRCA*2 families and the risk of skin cancer. Fam Cancer 2010; 9:489-93.

#### Glimm et al 2010

Glimm, E., Maurer, W., and Bretz, F. Hierarchical testing of multiple endpoints in group-sequential trials. Statistics in Medicine 2010;29, 219–228.

## Goodwin et al 2012

Goodwin PJ, Phillips KA, West DW, et al. Breast cancer prognosis in *BRCA*1 and *BRCA*2 mutation carriers: An international perspective breast cancer family registry population-based cohort study. J Clin Oncol 2012;30:19-26.

## Gupta et al 2007

Gupta B, Sait SN, Block AW, Ford LA, moysich KB, Baer MR. Acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) following treatment for ovarian cancer. J Clin Oncol 2007;ASCO Annual Meeting Proceedings Part 1,Vol 25, No 18S:17506.

## Hay et al 2009

Hay T, Matthews JR, Pietzka L, Lau A, Cranston A, Nygren AO, et al. Poly(ADP-ribose) polymerase-1 inhibitor treatment regresses autochthonous *BRCA* 2/p53-mutant mammary tumors in vivo and delays tumor relapse in combination with carboplatin. Cancer Res. 2009;69(9):3850-5.

# Helleday 2011

Helleday T. The underlying mechanism for the PARP and *BRCA* synthetic lethality: Clearing up the misunderstandings. Molecular Oncology 2011; 5: 387-393.

#### Hershman et al 2007

Hershman D, Neugut AI, Jacobson JS, Wang J, Tsai W, McBride R, Bennett CL, Grann VR. Acute Myeloid Leukemia or Myelodysplastic Syndrome Following Use of Granulocyte Colony-Stimulating Factors During Breast Cancer Adjuvant Chemotherapy. JNCI 2007 Vol. 99, Issue 3,Febr7.

## Honrado et al 2006

Honrado E, Benítez J, Palacios J. Histopathology of *BRCA1*- and *BRCA2*-associated breast cancer. Crit Rev Oncol Hematol. 2006;59:27-39

#### Hudis et al 2007

Hudis CA, William E, Barlow JP, Costantino RJ, Gray KI, Pritchard J-AW, et al. Proposal for Standardized Definitions for Efficacy End Points in Adjuvant Breast Cancer Trials: The STEEP System. J Clin Oncol 2007;25(15):2127-32.

## Huzarski et al 2013

Huzarski T, Byrski T et al. Ten-Year Survival in Patients With *BRCA*1-Negative and *BRCA*1-Positive Breast Cancer. J Clin Oncol 2013; 31:3191-3196.

#### Jeruss et al 2008

Jeruss SJ, Mittendorf EA et al. Combined Use of Clinical and Pathologic Staging Variables to Define Outcomes for Breast Cancer Patients Treated With Neoadjuvant Therapy. J Clin Oncol 2008; J Clin Oncol 26:246-252.

## Khatcheressian et al 2012

Khatcheressian JL, Hurley P et al. Breast Cancer Follow-Up and Management after primary treatment: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol 30, 2012.

### Kaufman et al 2014

Kaufman B, Shapira-Frommer R et al. Olaparib monotherapy in patients with advanced cancer and a germline *BRCA1/2* mutation. J Clin Oncol 2014 Nov 3. pii: JCO.2014.56.2728.

## Lachin 2005

Lachin, J. M. (2005). A review of methods for futility stopping based on conditional power. Statist. Med., 24: 2747–2764. Statist Med 24:2747-2764

## Liedtke et al 2008

Liedtke, C, Mazouni C, Hess K, Andre' F, Tordai A, Mejia JA, et al. Response to Neoadjuvant Therapy and Long-Term Survival in Patients With Triple-Negative Breast Cancer. Journal of Clinical Oncology; 2008 vol 26 no 8.

## Mavaddat et al 2012

Mavaddat et al. Pathology of breast and ovarian cancers among *BRCA*1 and *BRCA*2 mutation carriers: results from the Consortium of Investigators of Modifiers of *BRCA*1/2 (CIMBA)

Cancer Epidemiol Biomarkers Prev. 2012 January; 21(1): 134–147. doi:10.1158/1055-9965.EPI-11-0775.

## Metzger-Filho et al 2010

Metzger-Filho O, Tutt A, de Azambuja E, Saini KS, Viale G, Loi S, et al. Disecting the heterogeneity of triple negative breast cancer. J Clin Oncol. 2012 May 20;30 915:1879-87. Doi: 10.1200/JCO.2011.38.2010.

## Mieog et al 2007

Mieog JS, van der Hage JA, van de Velde CJ. Preoperative chemotherapy for women with operable breast cancer. Cochrane Database Syst Rev. 2007;18(2):CD005002.

#### Mittendorf et al 2011

Mittendorf EA, Jeruss JS, Tucker SL, Kolli A, Newman LA, Gonzalez-Angulo et al. Validation of a Novel Staging System for Disease-Specific Survival in Patients With Breast Cancer Treated With Neoadjuvant Chemotherapy. Journal of Clinical Oncology 2011 vol 29 no 15 may.

## Morton et al 2013

Morton LM, Dores GM, Tucker MA, Kim CJ, Onel K, Gilbert ES, et al. Evolving risk of therapy-related acute myeloid leukemia following cancer chemotherapy among adults in the United States, 1975-2008. Blood 2013;121(15):2996-3004.

## Murai et al 2012

Murai J, Huang SN, Das BB, Renaud A, et al. Trapping of PARP1 and PARP2 by Clinical PARP Inhibitors. AACR 2012; 72(21); 5588–99.

## Nardone et al (2015)

Nardone A, Goldstein A, Shea MJ, Mithchell T, Fu X, De C et al. PARP inhibition effects on endocrine therapy and resistance in estrogen receptor positive (ER+) breast cancer models. AACR 2015, abstract # 15LB8846AACR

## Praga et al 2005

Praga C, Bergh J, Bliss J, Bonneterre J, Cesana B, Coombes RC, et al. Risk of Acute Myeloid Leukemia and Myelodysplastic Syndrome in Trials of Adjuvant Epirubicin for Early Breast Cancer: Correlation With Doses of Epirubicin and Cyclophosphamide. Journal of Clinical Oncology 2005 Vol23 no 18 June.

## Rennert et al 2007

Rennert G, Bisland-Naggan S, Barnett-Griness O, Bar-Joseph N, Zhang S, Hedy S. Clinical outcomes of breast cancer in carriers of *BRCA*1 and *BRCA*2 mutations. N Engl J Med 2007;357:115-23.

## Rottenberg et al 2008

Rottenberg S, Jaspers JE, Kersbergen A, van der Burg E, Nygren AO, Zander SA, et al. High sensitivity of *BRCA*1-deficient mammary tumors to the PARP inhibitor AZD2281 alone and in combination with platinum drugs. Proc Natl Acad Sci. 2008;105(44):17079-84.

#### Robins et al 1991

Robins JM, Tsiatis AA. Correcting for noncompliance in randomized trials using rank preserving structural failure time models. Communications in Statistics - Theory and Methods 1991; 20:2609-2631.

#### Robson et al 2004

Robson ME, Chappuis PO, Satagopan J, Wong N, Boyd J, Goffin JR, et al. A combined analysis of outcome following breast cancer: Differences in survival based on *BRCA1/BRCA2* mutation status and administration of adjuvant treatment. Breast Cancer Res 2004;6(1):R8-17.

#### Robson et al 2017

Robson M, Im SA, Senkus E, Xu B, Domchek SM, Masuda N, et al. Olaparib for metastatic breast cancer in patients with a germline BRCA mutation. N Engl J Med 2017;377(6):522-33.

#### Schiewer et al 2013

Schiewer MJ, Goodwin JF, Han S, Brenner JC, Augello MA, Dean JL, et al. Dual roles of PARP-1 promote cancer growth and progression. Cancer Discov. 2012;2(12):1134-49

## Smith et al 2003

Smith RE, Bryant J, DeCillis A, Anderson S. Acute Myeloid Leukemia and Myelodysplastic Syndrome After Doxorubicin-Cyclophosphamide Adjuvant Therapy for Operable Breast Cancer: The National Surgical Adjuvant Breast and Bowel Project Experience 2003 J Clin Oncol 21:1195-1204.

## **Stone 2010**

A Stone. The application of bespoke spending functions in group-sequential designs and the effect of delayed treatment switching in survival trials. Pharmaceutical statistics 2010; 9, 151-161.

# Swain et al 2013

Swain SM, Tang G, Geyer CE Jr, Rastogi P, Atkins JN, Donnellan PP, et al. Definitive results of a phase III adjuvant trial comparing three chemotherapy regimens in women with operable, node-positive breast cancer: the NSABP B-38 trial. J Clin Oncol. 2013 Sep 10;31(26):3197-204.

#### Tryggvadottir et al 2013

Tryggvadottir L, Olafsdottir EJ, Olafsdottir GH, Sigurdsson H, Johannsson OT, Bjorgvinsson E, et al. Tumour diploidy and survival in breast cancer patients with BRCA2 mutations. Breast Cancer Res Treat 2013 Jul;140:375–38

#### Tutt et al 2010

Tutt A, Robson M, Garber JE, Domchek SM, Audeh MW, Weitzel JN, et al. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with *BRCA*1 or *BRCA*2 mutations and advanced breast cancer: a proof-of-concept trial. Lancet 2010; 376: 235–44.

## Vay et al 2011

Vay A, Kumar S, Seward S, Semaan A, Schiffer CA, Munkarah AR at al. Therapy-related myeloid leukemia after treatment for epithelial ovarian carcinoma: an epidemiological analysis. Gynecologic Oncology 2011;123:456-60.

#### Von Minckwitz et al 2012

Von Minckwitz G, Untch M, Blohmer JU et al. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol 2012; 30: 1796–1804.

#### Wesolowski et al 2007

Wesolowski R, Choueiri TK, Rybicki L, Shealy AG, Casey G, Weng D, et al. *BRCA* mutation status and risk of secondary malignancy following chemotherapy for breast cancer. J Clin Oncol, 2007;ASCO Annual Meeting Proceedings Part I. Vol (25);No. 18S (June 20 Supplement):11017.

## Yellen et al 1997

Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage 1997; 13(2), 63-74.

#### Zhang et al 2013

Zhang F, Wang Y, Wang L, Luo X, Huang K, Wang C, Du M, Liu F, Luo T, Huang D, Huang K. Poly(ADP-ribose) polymerase 1 is a key regulator of estrogen receptor α-dependent gene transcription. J Biol Chem. 2013;288(16):11348-57.

Clinical Study Protocol Appendix A Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5

Date 18 May 2018

#### Appendix A **Additional Safety Information**

## Further Guidance on the Definition of a Serious Adverse Event (SAE)

## Life threatening

'Life-threatening' means that the subject was at immediate risk of death from the AE as it occurred or it is suspected that use or continued use of the product would result in the subject's death. 'Life-threatening' does not mean that had an AE occurred in a more severe form it might have caused death (e.g., hepatitis that resolved without hepatic failure).

## Hospitalisation

Outsubject treatment in an emergency room is not in itself a serious AE, although the reasons for it may be (e.g., bronchospasm, laryngeal oedema). Hospital admissions and/or surgical operations planned before or during a study are not considered AEs if the illness or disease existed before the subject was enrolled in the study, provided that it did not deteriorate in an unexpected way during the study.

# Important medical event or medical intervention

Medical and scientific judgement should be exercised in deciding whether a case is serious in situations where important medical events may not be immediately life threatening or result in death, hospitalisation, disability or incapacity but may jeopardize the subject or may require medical intervention to prevent one or more outcomes listed in the definition of serious. These should usually be considered as serious.

Simply stopping the suspect drug does not mean that it is an important medical event; medical judgement must be used.

Examples of such events are:

- Angioedema not severe enough to require intubation but requiring iv hydrocortisone treatment
- Hepatotoxicity caused by paracetamol (acetaminophen) overdose requiring treatment with N-acetylcysteine
- Intensive treatment in an emergency room or at home for allergic bronchospasm
- Blood dyscrasias (e.g., neutropenia or anaemia requiring blood transfusion, etc.) or convulsions that do not result in hospitalisation
- Development of drug dependency or drug abuse

## A Guide to Interpreting the Causality Question

The following factors should be considered when deciding if there is a "reasonable possibility" that an AE may have been caused by the drug.

- Time Course. Exposure to suspect drug. Has the subject actually received the suspect drug? Did the AE occur in a reasonable temporal relationship to the administration of the suspect drug?
- Consistency with known drug profile. Was the AE consistent with the previous knowledge of the suspect drug (pharmacology and toxicology) or drugs of the same pharmacological class? OR could the AE be anticipated from its pharmacological properties?
- Dechallenge experience. Did the AE resolve or improve on stopping or reducing the dose of the suspect drug?
- No alternative cause. The AE cannot be reasonably explained by another aetiology such as the underlying disease, other drugs, other host or environmental factors.
- Rechallenge experience. Did the AE reoccur if the suspected drug was reintroduced after having been stopped? AstraZeneca would not normally recommend or support a rechallenge.
- Laboratory tests. A specific laboratory investigation (if performed) has confirmed the relationship?

A "reasonable possibility" could be considered to exist for an AE where one or more of these factors exist.

In contrast, there would not be a "reasonable possibility" of causality if none of the above criteria apply or where there is evidence of exposure and a reasonable time course but any dechallenge (if performed) is negative or ambiguous or there is another more likely cause of the AE.

In difficult cases, other factors could be considered such as:

- Is this a recognised feature of overdose of the drug?
- Is there a known mechanism?

Ambiguous cases should be considered as being a "reasonable possibility" of a causal relationship unless further evidence becomes available to refute this. Causal relationship in cases where the disease under study has deteriorated due to lack of effect should be classified as no reasonable possibility.

# Appendix B International Airline Transportation Association (IATA) 6.2 Guidance Document

# Labelling and shipment of biohazard samples

International Airline Transportation Association (IATA) classifies biohazardous agents into 3 categories. For transport purposes the classification of infectious substances according to risk groups was removed from the Dangerous Goods Regulations (DGR) in the 46th edition (2005). Infectious substances are now classified either as Category A, Category B or Exempt. There is no direct relationship between Risk Groups and categories A and B.

Category A Infectious Substances are infectious substances in a form that, when exposure to it occurs, is capable of causing permanent disability, life-threatening or fatal disease in otherwise healthy humans or animals. Category A pathogens are e.g., Ebola, Lassa fever virus:

• are to be packed and shipped in accordance with IATA Instruction 602.

**Category B Infectious Substances** are infectious Substances that do not meet the criteria for inclusion in Category A. Category B pathogens are e.g., Hepatitis A, B, C, D, and E viruses, Human immunodeficiency virus (HIV) types 1 and 2. They are assigned the following UN number and proper shipping name:

- UN 3373 Biological Substance, Category B
- are to be packed in accordance with UN3373 and IATA 650

**Exempt** - all other materials with minimal risk of containing pathogens

- Clinical trial samples will fall into Category B or exempt under IATA regulations
- Clinical trial samples will routinely be packed and transported at ambient temperature in IATA 650 compliant packaging
- Biological samples transported in dry ice require additional dangerous goods specification for the dry-ice content
- IATA compliant courier and packaging materials should be used for packing and transportation and packing should be done by an IATA certified person, as applicable
- Samples routinely transported by road or rail are subject to local regulations which require that they are also packed and transported in a safe and appropriate way to contain any risk of infection or contamination by using approved couriers and packaging / containment materials at all times. The IATA 650 biological sample containment standards are encouraged wherever possible when road or rail transport is used.

Clinical Study Protocol Appendix C Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5









Clinical Study Protocol Appendix D Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5

Date 18 May 2018

#### **Appendix D Actions Required in Cases of Increases in Liver** Biochemistry and Evaluation of Hy's Law

## Introduction

This Appendix describes the process to be followed in order to identify and appropriately report cases of Hy's Law. It is not intended to be a comprehensive guide to the management of elevated liver biochemistries.

During the course of the study the Investigator will remain vigilant for increases in liver biochemistry. The Investigator is responsible for determining whether a subject meets potential Hy's Law (PHL) criteria at any point during the study.

The Investigator participates, together with AstraZeneca clinical project representatives, in review and assessment of cases meeting PHL criteria to agree whether Hy's Law (HL) criteria are met. HL criteria are met if there is no alternative explanation for the elevations in liver biochemistry other than Drug Induced Liver Injury (DILI) caused by the Investigational Medicinal Product (IP).

The Investigator is responsible for recording data pertaining to PHL/HL cases and for reporting Adverse Events (AE) and Serious Adverse Events (SAE) according to the outcome of the review and assessment in line with standard safety reporting processes.

#### **Definitions**

# Potential Hy's Law (PHL)

Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)  $\geq 3x$  Upper Limit of Normal (ULN) together with Total Bilirubin (TBL)  $\geq 2xULN$  at any point during the study following the start of study medication irrespective of an increase in Alkaline Phosphatase (ALP).

## Hy's Law (HL)

AST or ALT  $\geq 3x$  ULN **together with** TBL  $\geq 2x$ ULN, where no other reason, other than the IMP, can be found to explain the combination of increases, e.g., elevated ALP indicating cholestasis, viral hepatitis, another drug.

For PHL and HL the elevation in transaminases must precede or be coincident with (i.e. on the same day) the elevation in TBL, but there is no specified timeframe within which the elevations in transaminases and TBL must occur.

# **Identification of Potential Hy's Law Cases**

In order to identify cases of PHL it is important to perform a comprehensive review of laboratory data for any subject who meets any of the following identification criteria in isolation or in combination:

- ALT  $\geq 3$ xULN
- AST  $\geq 3xULN$
- TBL  $\geq 2xULN$

The Investigator will without delay review each new laboratory report and if the identification criteria are met will:

- Determine whether the subject meets PHL criteria (see Section Definitions within this Appendix for definition) by reviewing laboratory reports from all previous visits
- Promptly enter the laboratory data into the laboratory CRF

# Follow-up

## Potential Hy's Law Criteria not met

If the subject does not meet PHL criteria the Investigator will:

 Perform follow-up on subsequent laboratory results according to the guidance provided in the Clinical Study Protocol.

# Potential Hy's Law Criteria met

If the subject does meet PHL criteria the Investigator will:

Notify the AstraZeneca representative who will then inform the central Study Team

The Study Physician contacts the Investigator, to provide guidance, discuss and agree an approach for the study subjects' follow-up and the continuous review of data. Subsequent to this contact the Investigator will:

- Monitor the subject until liver biochemistry parameters and appropriate clinical symptoms and signs return to normal or baseline levels, or as long as medically indicated.
- Investigate the etiology of the event and perform diagnostic investigations as discussed with the Study Physician.
- Complete the three Liver CRF Modules as information becomes available.
- If at any time (in consultation with the Study Physician) the PHL case meets serious criteria, report it as an SAE using standard reporting procedures.

# Review and Assessment of Potential Hy's Law Cases

The instructions in this Section should be followed for all cases where PHL criteria are met.

No later than 3 weeks after the biochemistry abnormality was initially detected, the Study Physician contacts the Investigator in order to review available data and agree on whether there is an alternative explanation for meeting PHL criteria other than DILI caused by the IMP. The AstraZeneca Medical Science Director and Global Safety Physician will also be involved in this review together with other subject matter experts as appropriate.

According to the outcome of the review and assessment, the Investigator will follow the instructions below.

If there is an agreed alternative explanation for the ALT or AST and TBL elevations, a determination of whether the alternative explanation is an AE will be made and subsequently whether the AE meets the criteria for a SAE:

- If the alternative explanation is **not** an AE, record the alternative explanation on the appropriate CRF
- If the alternative explanation is an AE/SAE, record the AE /SAE in the CRF accordingly and follow the AZ standard processes

If it is agreed that there is **no** explanation that would explain the ALT or AST and TBL elevations other than the IMP:

- Report an SAE (report term 'Hy's Law') according to AstraZeneca standard processes.
  - The 'Medically Important' serious criterion should be used if no other serious criteria apply
  - As there is no alternative explanation for the HL case, a causality assessment of 'related' should be assigned.

If, there is an unavoidable delay, of over 3 weeks, in obtaining the information necessary to assess whether or not the case meets the criteria for HL, then it is assumed that there is no alternative explanation until such time as an informed decision can be made:

- Report an SAE (report term 'Potential Hy's Law') applying serious criteria and causality assessment as per above
- Continue follow-up and review according to agreed plan. Once the necessary supplementary information is obtained, repeat the review and assessment to determine whether HL criteria are met. Update the SAE report according to the outcome of the

review amending the reported term if an alternative explanation for the liver biochemistry elevations is determined.

# Actions Required for Repeat Episodes of Potential Hy's Law

This section is applicable when a subject meets PHL criteria on study treatment and has already met PHL criteria at a previous on study treatment visit.

The requirement to conduct follow-up, review and assessment of a repeat occurrence(s) of PHL is based on the nature of the alternative cause identified for the previous occurrence.

The investigator should determine the cause for the previous occurrence of PHL criteria being met and answer the following question:

• Was the alternative cause for the previous occurrence of PHL criteria being met found to be the disease under study e.g. chronic or progressing malignant disease, severe infection or liver disease?

If No: follow the process described in Potential Hy's Law Criteria met of this Appendix

#### If Yes:

Determine if there has been a significant change in the subject's condition<sup>#</sup> compared with when PHL criteria were previously met

- If there is no significant change no action is required
- If there is a significant change follow the process described in Section Follow-up of this Appendix

<sup>#</sup> A 'significant' change in the subject's condition refers to a clinically relevant change in any of the individual liver biochemistry parameters (ALT, AST or total bilirubin) in isolation or in combination, or a clinically relevant change in associated symptoms. The determination of whether there has been a significant change will be at the discretion of the Investigator; this may be in consultation with the Study Physician if there is any uncertainty.

#### References

FDA Guidance for Industry (issued July 2009) 'Drug-induced liver injury: Premarketing clinical evaluation'

# **Appendix E** Acceptable Birth Control Methods

# Olaparib is regarded as a compound with medium/high foetal risk.

Women of childbearing potential and their partners, who are sexually active, must agree to the use of TWO highly effective forms of contraception in combination (as listed below). This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug, or they must totally/truly abstain from any form of sexual intercourse (see below).

Male patients must use a condom during study treatment and for 3 months after last dose of study drug when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Male patients should not donate sperm throughout the period of taking study treatment and for 3 months following the last dose of study drug.

## Acceptable Non-hormonal birth control methods include

- Total/True abstinence: When the patient refrains from any form of sexual intercourse and this is in line with their usual and/or preferred lifestyle, this must continue for the total duration of the treatment period and for 1 month after the last dose of study drug for female patients, for 3 months after last dose for male patients. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods, or declaration of abstinence solely for the duration of a trial) and withdrawal are not acceptable methods of contraception]
- Vasectomised sexual partner plus male condom. With participant assurance that partner received post-vasectomy confirmation of azoospermia
- Tubal occlusion plus male condom
- IUD plus male condom. Provided coils are copper-banded

## Acceptable hormonal methods

- Etonogestrel implants (e.g., Implanon, Norplan) PLUS male condom
- Normal and low dose combined oral pills PLUS male condom
- Norelgestromin / EE transdermal system PLUS male condom
- Intravaginal device (e.g., EE and etonogestrel) PLUS male condom
- Cerazette (desogestrel) PLUS male condom. Cerazette is currently the only highly efficacious progesterone based pill.
- Hormonal shot or injection (e.g., Depo-Provera) PLUS male condom

• Intrauterine system [IUS] device (e.g., levonorgestrel releasing IUS -Mirena®) PLUS male condom

#### Appendix F **ECOG Performance Status**

# **Example of Performance Status (ECOG SCALE)**

| DESCRIPTION | ECOG GRADE |
|---|---|
| Fully active, able to carry on all pre-disease performance without restriction. | 0 |
| Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, i.e. light housework, office work. | 1 |
| Ambulatory and capable of self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. | 2 |
| Capable of only limited self care, confined to bed or chair more than 50% of waking hours. | 3 |
| Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. | 4 |

# **Appendix G** Patient Reported Outcomes (FACIT-Fatigue, EORTC QLQ-C30)

# FACIT Fatigue Scale (Version 4)

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the <u>past 7 days</u>.

| | | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very |
|---|---|---|---|---|---|---|
| an) | I feel fatigued | U | 1 | 2 | 3 - | 4 |
| HIII | I feel weak all over | 0 | 1 | 2 | 3 | 4 |
| Ast | I feel listless ("washed out") | 0 | 1 | 2 | 3 | 4 |
| AaZ | 1 feel tired | 0 | 1 | 2 | 3 | 4 |
| A163 | I have trouble starting things because I am tired | 0 | 1 | 2 | 3 | 4 |
| Anv | I have trouble finishing things because I am tired | 0 | 1 | 2 | 3 | 4 |
| Ans | 1 have energy | 0 | 1 | -2 | 3 | 4 |
| An7 | I am able to do my usual activities | 0. | 1 | 2 | 3 | 4 |
| Asir | I need to sleep during the day | 0 | 1 | 2 | 3 | 4 |
| Aut2 | I am too tired to eat | 0 | 1 | 2 | 3 | 4 |
| Anis | I need help doing my usual activities | 0 | 1 | 2 | 3 | 4 |
| Asid | I am frustrated by being too tired to do the things I want to do | 0 | 1 | 2 | 3 | 4 |
| Anti- | I have to limit my social activity because I am tired | Ω | 1 | 2 | 3 | 4 |

 Biglids (Driversal)
 14 Ministrator

 Copyright 1997, 1997
 "Ress Is

Clinical Study Protocol Appendix G Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5

Date 18 May 2018



# EORTC QLQ-C30 (version 3)

Please fill in your initials:

We are interested in some things about you and your health. Please answer all of the questions yourself by circling the number that best applies to you. There are no "right" or "wrong" answers. The information that you provide will remain strictly confidential.

| | ar birthdate (Day, Month, Year): lay's date (Day, Month, Year): 31 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | | | |
|---|---|---|---|---|---|
| | 1) | Not at | A<br>Little | Quite<br>a Bit | Very<br>Much |
| 1. | Do you have any trouble doing strenuous activities,<br>like carrying a heavy shop ing bag or a suitcase? | 1 | 2 | 3 | 4 |
| 2, | Do you have any trouble taking a long walk? | 1 | 2 | 3 | 4 |
| 3. | Do you have any trouble taking a short walk outside of the house? | Í | 2 | 3 | 4 |
| 4. | Do you need to stay in bed or a chair during the day? | 1 | 2 | 3 | 4 |
| 5. | Do you need help with eating, dressing, washing yourself or using the toilet? | 1 | 2 | 3 | 4 |
| Du | ring the past week: | Not at | A<br>Little | Quite<br>a Bit | Very<br>Much |
| 6. | Were you limited in doing either your work or other daily activities? | -)1 | 2 | 3 | 4 |
| 7. | Were you limited in pursuing your hobbies or other leisure time activities? | 1 | 2 | 3 | 4 |
| 8. | Were you short of breath? | 1 | -2) | 3 | 4 |
| 9. | Have you had pain? | 1 | 1/2 | 3 | 4 |
| 10. | Did you need to rest? | | 2 | 1 | 4 |
| 11. | Have you had trouble sleeping? | -1 | 1 | 3 | 4 |
| 12. | Have you felt weak? | 1 | 2 | 3 | 4 |
| 13, | Have you lacked appetite? | 1 | 12 | 3 | 4 |
| 14. | Have you felt nauseated? | 1 | 2 | 3 | 4 |
| 15. | Have you vomited? | 1 | 2 | 3 | 4 |
| 16. | Have you been constipated? | 1 | 2 | 3 | 4 |

Please go on to the next page

Clinical Study Protocol Appendix G Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5

| | | - | |
|------|----|-----|------|
| Date | 18 | May | 2018 |

| During the past week: | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|
| 17. Have you had diarrhea? | 1 | 2 | 3 | 4 |
| 18. Were you tired? | 1 | 2 | 3 | 4 |
| 19. Did pain interfere with your daily activities? | 1 | 2 | 3 | 4 |
| 20. Have you had difficulty in concentrating on things,<br>like reading a newspaper or watching television? | í | 2 | 3 | 4 |
| 21. Did you feel tense? | 1 | 2 | 3 | 4 |
| 22. Did you worry? | 1 | 2 | 3 | 4 |
| 23. Did you feel irritable? | 1 | 2 | 3 | 4 |
| 24. Did you feel depressed? | 1 | 2 | 3 | 4 |
| 25. Have you had difficulty remembering things? | 1 | 2 | 3 | 4 |
| 26. Has your physical condition or medical treatment interfered with your family life? | 1 | 2 | 3 | 4 |
| Has your physical condition or medical treatment interfered with your <u>social</u> activities? | 1 | 2 | 3 | 4 |
| 28. Has your physical condition or medical treatment caused you financial difficulties? | Í | 2 | 3 | 4 |
| For the following questions please circle the number best applies to you 29. How would you rate your overall health during the past week? | betwe | en 1 a | nd 7 1 | that |
| 1 2 3 4 5 6 | 4 | 1 | | |
| | cellent | / | <u>()</u> | |
| 30. How would you rate your overall quality of life during the past week? | | | / | |
| 1 2 3 4 5 6 | 7 | | | |
| Very poor Ex | cellent | | | |

 $\ \, \ \, \ \,$  Copyright 1995 EORTC Quality of Life Group. All rights reserved, Version 3.0



Clinical Study Protocol Appendix #H Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Version 5

Date 18 May 2018

#### **CPS & EG score Appendix H**

Calculation instructions: Add the points for Clinical Stage + Pathologic Stage + ER status + Nuclear grade to derive a sum (CPS&EG score) between 0 and 6.

Table 18 Point assignments for the CPS + EG staging system

| Stag | e/feature | Points |
|---|---|---|
| | I | 0 |
| | IIA | 0 |
| Clinical Stage | IIB | 1 |
| (AJCC staging <sup>1</sup> ) | IIIA | 1 |
| | IIIB | 2 |
| | IIIC | 2 |
| | 0 | 0 |
| | I | 0 |
| | IIA | 1 |
| Pathologic Stage (AJCC staging <sup>1</sup> ) | IIB | 1 |
| (risee staging) | IIIA | 1 |
| | IIIB | 1 |
| | IIIC | 2 |
| Receptor status | ER negative <sup>2</sup> | 1 |
| Nuclear grade <sup>3</sup> | Nuclear grade 3 | 1 |

AJCC: American Joint Committee on Cancer (https://cancerstaging.org/Pages/default.aspx).

ER: Estrogen receptor; definitions for ER negativity see eligibility criteria Section 4.1.4.a.

In the unlikely situation nuclear grade cannot be determined, regular histologic grade should be used; if only Nottingham overall grade is reported, the Nottingham overall grade must be 9 to be scored as 1 point in the CPS&EG score (http://pathology.jhu.edu/breast/grade.php).

# **SIGNATURE PAGE**

This is a representation of an electronic record that was signed electronically and this page is the manifestation of the electronic signature

| Document Name: d081cc00006-csp-v5-clean | | |
|---|---|---|
| <b>Document Title:</b> | D081CC00006 Clinical Study Protocol Version 5 Clean | |
| Document ID: | Doc ID-003797115 | |
| Version Label: | 1.0 CURRENT LATEST APPROVED | |
| Server Date<br>(dd-MMM-yyyy HH:mm 'UTC'Z) | Signed by Meaning of Signature | |
| 21-May-2018 16:33 UTC | | Author Approval |
| 21-May-2018 15:51 UTC | Author Approval | |
| 21-May-2018 14:51 UTC | Author Approval | |
| 21-May-2018 14:22 UTC | | Content Approval |

Notes: (1) Document details as stored in ANGEL, an AstraZeneca document management system.

## **SUMMARY OF CHANGES - PROTOCOL**

For Protocol Amendment #7 to: NSABP B-55/BIG 6-13

NCI Protocol #: NSABP B-55

Local Protocol #: NSABP B-55/BIG 6-13

NCI Version Date: 05/06/2021

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | NSABP PROTOCOL<br>B-55/BIG 6-13 | 2 | Amendment 7 was added to the Document History table with a Version Date of May 6, 2021. |

The following sections of the protocol were revised to clarify AE/SAE reporting requirements. This amendment is necessary to align the reporting requirements for second primary malignancies between the U.S. and the Rest of World versions of the protocol. Protocol text was revised as necessary to delete instructions differentiating reporting instructions for treatment-related secondary malignancies and non-treatment related second malignancies. Clarifications were also made for the reporting of non-melanoma skin cancers and carcinoma in situ cases as non-serious AEs, irrespective of the timing of the event in relation to study therapy, unless one of the criteria for seriousness is met.

| | the event in relation to study therapy, timess one of the criteria for seriousness is met. | | |
|---|---|---|---|
| 2. | 3.1<br>Table 3 | 54 | Footnote e was revised. |
| 3. | 6.4.8.2 | 101 | Information from the Secondary malignancy section was moved to Section 6.4.8.2 to consolidate information. Treatment-related secondary malignancies and non-treatment related second malignancies are not being differentiated for reporting purposes. |
| 4. | 6.4.9 Time period for collection of adverse events | 103 | Paragraph 2 was revised. |
| 5. | 6.4.9<br>Adverse events after<br>the 30-day follow up<br>period | 104 | Paragraph 1 was revised. |
| 6. | 6.4.9<br>Secondary<br>malignancy | 107 | Instructions for reporting secondary malignancies was moved from the Secondary malignancy section was moved to Section 6.4.8.2. |
| 7. | 6.4.9<br>New cancers | 108 | Paragraph 1 was revised. Paragraph 2 was deleted because the information can be found in Section 6.4.8.2. |
| 8. | 6.4.9<br>Olaparib adverse<br>events of special<br>interest | 109 | Paragraph 1 was revised. |

# **SUMMARY OF CHANGES - PROTOCOL**

For Protocol Amendment #6 to: NSABP B-55/BIG 6-13

NCI Protocol #: NSABP B-55

Local Protocol #: NSABP B-55/BIG 6-13

NCI Version Date: 07/27/18

Protocol Title: A Randomised, Double-Blind, Parallel Group, Placebo-Controlled Multi-Centre Phase III Study to Assess the Efficacy and Safety of Olaparib Versus Placebo as Adjuvant Treatment in Patients with Germline BRCA1/2 Mutations and High Risk HER2 Negative Primary Breast Cancer Who Have Completed Definitive Local Treatment and Neoadjuvant or Adjuvant Chemotherapy

The primary reason for this protocol amendment is to revise the sample size of the study. In addition, revisions have been made to align with current practice, safety updates, and to clarify procedures. Minor editorial changes have also been made but are not included in this summary table.

#### **Statistical background - Rationale for amendment:**

To support the addition of the ER-positive cohort in Amendment 2, a simulation study was undertaken with the objective to predict accrual of events and, therefore, the timing of the interim and primary analyses. The simulation study included relevant operating characteristics for the anticipated possible proportions enrolled in each of the 4 subgroups, survival was modelled by piecewise exponential distribution for which annualised hazard according to the respective subgroups were taken from the most recent published data (Dent et al 2007, Cortazar et al 2014, Swain et al 2013).

Following the observation of lower than anticipated event rate (using data extracted on 25 August 2017), it was clear that the published data used for the simulations were too pessimistic with respect to event rates for the triple-negative adjuvant population that have been recruited into Study D081CC00006 (OlympiA) since 2014.

Further predictions were run using the current data (extract date 10 November 2017) and applying AstraZeneca's 'Shiny' oncology event prediction R package. A survival model assuming a Weibull distribution was fitted to the previous study data and used to predict future survival times. Whilst the simulation study simulated over varying proportions enrolled in each subgroup, by using the current data, the predictions were based on 1153 patients of whom 15% were ER-positive and the ratio of Adjuvant to Neoadjuvant was roughly 1:1. An 8% drop-out rate for the first 12 months, not previously included, was incorporated based on the rate observed so far. The programme forecasted future enrolment from 1153 to 1800 based on the recent observed enrolment rate. There was also no need to adjust this forecast for delays in enrolment due to the protocol amendment.

Given the predictions for timing of the interim and primary analyses, it was decided to increase the sample size to 1800 and for the power to remain at 90%. Because the event rate was lower than anticipated, the restriction to have a minimum 2-year follow-up after the last patient enrolled could be removed. Patient enrolled continue about one year longer than originally anticipated and more patients would be enrolled, thus providing an increase in the number of patient years of follow-up at the time of primary analysis even without the 2-year minimum follow-up criterion.

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | NSABP PROTOCOL | 2 | Amendment 6 was added to the Document History table |
| | B-55/BIG 6-13 | | with a Version Date of July 27, 2018. |
| 2. | Title Page | 3 | Merck logo added to the Rest of World protocol Title page. |
| | | | Merck has joined with AstraZeneca in the co-development |
| | | | and co-commercialization of olaparib. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 3. | List of Olympia<br>Protocol Authors | 4-5 | The list of protocol authors has been updated. |
| 4. | List of Abbreviations<br>and Definition of<br>Terms | 23, 26,<br>27 | The following abbreviations and definition of terms were added: • AESI Adverse event of special interest • PFS2 Time to second progression • TPC Chemotherapy of physician's choice |
| 5. | Protocol Synopsis 3.2.3 12.2.3.2 12.2.7 | 6, 8, 12<br>56<br>143<br>149 | <ul> <li>The number of patients planned has been increased from 1500 to 1800.</li> <li>The number of centres participating in the study has increased from 500 to 700.</li> <li>The number of patients anticipated to be enrolled by the US was changed from 300 to 230 and the Rest of World was changed from 1200 to 1570.</li> </ul> |
| 6. | Protocol Synopsis<br>12.2.7 | 12<br>149 | The estimation of time for study recruitment has been increased to 5 years (previously 4 years) to account for the 300 additional patients. |
| 7. | Protocol Synopsis<br>6.2.5<br>12.2.1.1<br>12.2.2<br>12.2.7 | 12<br>98<br>136<br>139<br>149 | The text "minimum 24 month follow-up" was removed from the data cut-off for the primary analysis as the expected high event rate in the first 2 years has not been seen. |
| 8. | Protocol Synopsis<br>12.1.1<br>12.2.6 | 12<br>135<br>146 | Interim analysis will now be triggered by events in the first 900 patients (previously 750 patients). |
| 9. | 1.1.9.1 | 32 | Efficacy data for Study D0819C00003 (OlympiAD) was added to the background. |
| 10. | 1.4 | 39 | Information was added to the Potential benefit section about the olaparib tablet formulation approval for patients with deleterious or suspected deleterious <i>gBRCAm</i> , HER2-negative metastatic breast cancer. |
| 11. | 3.1, Figure 1, Table 1,<br>Table 2, Table 3<br>3.2.1<br>6.2.1<br>6.2.2<br>6.2.3<br>6.3.1 | 42, 44,<br>48, 49,<br>51, 53,<br>54, 55,<br>94, 97,<br>99 | The text regarding mammogram and/or breast MRI scans was amended to include ipsilateral and/or contralateral scanning. Clarification was provided regarding the use of ultrasound in patients who underwent a bilateral mastectomy and for male patients. |
| # | Section | Page(s) | Change |
|---|---|---|---|
| 12. | 3.1 Table 3 | 54 | Information was added to footnote e to clarify<br>monitoring of all ongoing AEs/SAEs and any new<br>AEs/SAEs identified during the 30 calendar days. |
| | | | <ul> <li>Pneumonitis was included in the events occurring after<br/>the 30 day follow-up period that should be reported as<br/>an SAE. New primary malignancy was revised to new<br/>treatment-related secondary malignancy to be<br/>consistent with CTEP terminology.</li> </ul> |
| 13. | 3.1 Table 1<br>3.1 Table 2<br>6.2.1<br>6.2.2<br>6.4.15.1 | 47<br>49, 51<br>94<br>96<br>114 | <ul> <li>Footnote i was revised to clarify instructions regarding a positive pregnancy test at baseline. Instructions for a positive pregnancy test during the study were deleted.</li> <li>Additional time points for pregnancy testing in women of childbearing potential were added to Table 2. The time points for pregnancy testing were added to align with the AstraZeneca Olaparib Standard Protocol 2018. Footnote a was revised to clarify instructions regarding</li> </ul> |
| | | | <ul> <li>a positive pregnancy test during the study.</li> <li>Pregnancy tests on blood or urine was changed to serum or urine for consistency throughout the protocol.</li> </ul> |
| 14. | 4.1 | 61-62 | Criterion 11B: The text describing methods of contraception was revised. |
| 15. | 4.2 | 63-64 | Criterion 11: The use of strong and moderate CYP3A inhibitors text was revised, and new criteria were included to cover the use of concomitant strong and moderate CYP3A inducers on study. |
| | | | <ul> <li>Criterion 13: Criteria were modified for patients with a<br/>current or past history of haematologic malignancies<br/>and any clonal non-malignant haematological disorder<br/>which predisposes the patient to develop a<br/>haematological malignancy.</li> </ul> |
| 16. | 5.1.1 | 64 | A new section was added to indicate that the consumption of grapefruit juice while on study is prohibited. |
| 17. | 5.1.2<br>Appendix E | 64-65<br>176 | Text was updated to specify that two highly effective forms of contraception should be used in combination, and this should be started from the signing of the informed consent to be consistent with the text in Appendix E. Male patient contraception text clarified. |
| 18. | 5.2.4 | 69 | Text was added to be consistent with CTSU template language for OPEN. |
| 19. | 5.5.2.1<br>5.5.12.2 | 72, 79<br>82 | <ul> <li>Table 5 and Table 6 were updated to include temporary dose reductions to 300 and 200 mg due to CYP3A inhibitor exposure.</li> <li>Table 8 and Table 9 were added to cover dose reductions for management of renal impairment and the use of strong or moderate CYP3A inhibitors while on study, respectively.</li> </ul> |

| # | Section | Page(s) | |
|---|---|---|---|
| 20. | 5.5.8 | 77 | The OAOP website address was updated to |
| | | | https://ctepcore.nci.nih.gov/OAOP. |
| 21. | 5.5.12.3 | 82 | A new section to cover management of renal impairment |
| | | | while on study was added. |
| 22. | 5.5.12.7 | 83-84 | <ul> <li>The recording of reasons for reductions/interruptions was clarified.</li> <li>The type of biopsy procedure for which no stoppage of study treatment is required was clarified.</li> <li>Additional text was provided advising caution while driving or using machinery in case of AEs of asthenia, fatigue and dizziness.</li> </ul> |
| 23. | 5.6.2 | 84-88 | <ul> <li>Section name was changed from CYP3A to Restricted concomitant medications.</li> <li>CYP3A text is now summarised in Table 10. Sections 5.6.3, 5.6.4, and 5.6.6 of the September 28, 2017, version of the protocol were deleted, and the information was included in Table 10.</li> </ul> |
| 24. | 6.2.1 | 95 | The capturing of adverse events during Screening text has been revised to reflect current practice. |
| 25. | 6.4.4 | 100 | CTCAE v4.0 will be used for AE reporting and CTCAE v5.0 will be used for SAE reporting. |
| 26. | 6.4.7 | 101 | Sore throat was deleted so that the list in Section 6.4.7 is reflective of the informed consent form. |
| 27. | 6.4.8.2 | 103 | Protocol-specific reporting requirements were revised to include pneumonitis. |
| 28. | 6.4.9 | 105-<br>106<br>107<br>110 | <ul> <li>The recording of adverse events text has been revised to reflect current practice.</li> <li>A section for recording of adverse events after the 30 day follow up period has been added.</li> <li>CTCAE grade and changes in CTCAE grade has been included in the list of variables collected for each AE.</li> <li>New cancers: Reporting of new primary cancers was clarified. Text was added to indicate that new primary cancers are considered as IDFS event and must be reported on the endpoint CRF. Patients with new primary cancers which require (neo)adjuvant treatment of any kind for appropriate management must be discontinued from study treatment.</li> <li>A new section for olaparib adverse events of special interest (AESI) was added. The AESIs are MDS/AML, new treatment-related secondary malignancy (other than MDS/AML), and pneumonitis.</li> <li>A questionnaire will be sent to any investigator</li> </ul> |
| | | | reporting an AESI as an aid to provide further detailed information on the event. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 29. | 3.1 Table 2 (footnote h) 6.8 | 51<br>121 | Text was included to clarify that samples should be collected preferably on visit 4, day 29; however, samples can also be taken at a later treatment visit, provided that PK consent was obtained beforehand. |
| 30. | 5.9<br>11.1.2.1 | 91<br>132 | Text regarding a survival sweep was deleted from the protocol. |
| 31. | 12.2.1.1<br>12.2.7 | 136<br>149 | <ul> <li>Text was updated for the predicted timing of the primary analysis.</li> <li>Text relating to ER-positive cohorts was deleted as the revised predictions are based on the current data which has approximately 15% ER-positive patients.</li> </ul> |
| 32. | 12.2.1.2 | 137 | Details of sensitivity analyses were included where the results of ER and PgR status from the local and central labs differ in >5% of randomised patients. |
| 33. | 12.2.1.3<br>12.2.2 | 137<br>139 | Text was revised for number of events below which it is not considered appropriate to present analyses. |
| 34. | 12.2.3.2 | 143 | Patient reported outcomes sample size estimates were updated based on the sample size increase. |
| 35. | 12.2.6 | 146-<br>147 | Text for predicted timing of the interim analysis was updated. |
| 36. | 12.2.7 | 150-<br>151 | <ul> <li>Table 13 was replaced with a new version based on the actual accrual pattern between June 2014 and February 2018. The table has been renumbered to Table 16.</li> <li>Table 14 and text related to this table have been deleted.</li> </ul> |
| 37. | 12.2.8 Table 17 | 152 | Table was updated with new US accrual expectation of 230 patients. |
| 38. | 13.2 | 154 | Additional text concerning what constitutes an overdose has been added. |
| 39. | 13.3.2 | 155 | Fetal death was changed to pregnancy loss to match the CTCAE v5.0 term. |
| 40. | 14. | 163 | A new reference, Robson et al 2017, was included to support the new data added to Section 1.1.9.1. |
| 41. | Appendix H | | Appendix H from the September 28, 2017, version of the protocol was deleted as the text is now contained within Section 5.6.2. The subsequent appendix was relettered. |
| 42. | Appendix I | 185 | A typographical error in footnote 2 was corrected from 4.1.3a to 4.1.4a. Appendix relettered to Appendix H. |

For Protocol Amendment #5 to: NSABP B-55/BIG 6-13

NCI Protocol #: NSABP B-55

Local Protocol #: NSABP B-55/BIG 6-13

NCI Version Date: 09/28/17

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | NSABP<br>PROTOCOL<br>B-55/BIG 6-13 | 1 | Amendment 5 was added to the Document History table with a Version Date of September 28, 2017. |
| 2. | 5.2 | 62-66 | New CTSU language regarding the Registration and Credentialing Repository (RCR) was added to Sections 5.2.1, 5.2.2.1, 5.2.2.5, and 5.2.4, pages 62-66 as requested by CTEP. |
| 3. | 5.5.8 | 74 | As requested by CTEP, the PMB IB Coordinator e-mail was deleted from Section 5.5.8 because the instructions for obtaining a copy of the IB are located in Section 5.5.4. |
| 4. | 6.1.2 | 86-87 | New CTSU language for data submission via Medidata Rave was added. |
| 5. | 6.4.7 | 95 | Fever and sore throat were added to the list of common adverse events associated with olaparib based on changes in the Request for Rapid Amendment dated September 6, 2017. |

For Protocol Amendment #4 to: NSABP B-55/BIG 6-13

NCI Protocol #: NSABP B-55

Local Protocol #: NSABP B-55/BIG 6-13

NCI Version Date: 07/25/17

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | | | Multiple editorial changes were made to the protocol to correspond to changes made to the protocol version which covers all patients outside the United States (where AstraZeneca is the sponsor). The individual changes are not outlined in the Summary of Changes. |
| 2. | NSABP<br>PROTOCOL<br>B-55/BIG 6-13 | 1 | The Protocol Pathologist was changed from the protocol Pathologist was c |
| 3. | Clinical Study<br>Protocol | 2 | Version 4 and 23 March 2017 were added to document the current version and date of the protocol that covers all patients outside the United States (where AstraZeneca is the sponsor). The AstraZeneca Research and Development Representative information and amendment information were deleted by AstraZeneca. |
| • | | | |
| 5. | Table of Contents | 18-19 | The list of appendices was updated to reflect the deletion of Appendix A, and the relettering of subsequent appendices. |
| 6. | Information<br>Resources | 20<br>21 | Row 5, column 3: IRB approvals must be submitted to CTSU via the Regulatory Submission Portal. Row 2, column 3: The fax number for the SAE reporting nurse was changed from 412-622-2113 to 412-624-1082. |
| 7. | Cancer Trials Support Unit (CTSU) Address and Contact Information | 22-23 | The CTSU information table was updated to the current CTSU text for patient enrollment, data submission, and access to the CTSU website. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 8. | List of Abbreviations and Definition of Terms | 24,<br>25, 27 | <ul> <li>The following were deleted from the list: BIG Breast International Group non pCR Non-polymerase chain reaction</li> <li>ECOG was revised to include performance status and its definition.</li> <li>CTEP-IAM was moved to follow CTEP-AERS so the terms would be in alphabetical order.</li> </ul> |
| 9. | 1.3 | 35 | Paragraph 2: Inclusion criteria 3b, 5, 6 were renumbered to 3A, 3B, and 4b to be consistent with the protocol version which covers all patients outside the United States (where AstraZeneca is the sponsor). |
| 10. | Table 3 | 53 | Footnote a: The reference to bilateral mastectomy was deleted to match the text in Table 2, footnote e. |
| 11. | Inclusion criteria 4a and 4b | 57-58 | The requirement for TNBC that all ER and PgR assessments that are locally available must be negative text for determining ER status has been deleted from the July 25, 2017, version of the protocol. For ER and/or PgR positive patients, the text that any tumour that has been locally assessed as ER and/or PgR positive in either the core biopsy or the surgical specimen is considered to be ER and/or PgR positive. The text deleted from the July 25, 2017, protocol version had been added to the October 19, 2015, version of the protocol, but it was subsequently determined that the requirement was overly restrictive for patients with breast cancer tumours classified as triple-negative based on the receptor status analysis from the core needle biopsy but who had low levels of peroxidase staining for ER and PgR in their postneoadjuvant surgical specimen. For eligibility, the lesion considered at highest risk for recurrence based on the investigator's discretion will be used for eligibility determination. By deleting the text, the July 25, 2017, version of the protocol reverts to the July 22, 2014, version of the protocol. |
| 12. | 5.2.3.1<br>5.2.3.2<br>5.2.3.3<br>5.2.3.4<br>5.2.3.5 | 65-67 | Revised CTSU template text regarding IRB approval, site registration, and submission of regulatory documents was added to the current version of the protocol. |
| 13. | 5.5.5 | 74-75 | Paragraph 7: Revised template text from the NCI Pharmaceutical Management Branch (PMB) describing who may request NCI-supplied agents was added. |
| 14. | 5.5.7 | 75 | Revised template text from the NCI Pharmaceutical Branch describing the requirements for requesting CTEP-supplied investigational agents was added. |
| 15. | 5.5.8 | 75 | A list of useful PMB and CTEP links and contacts was added. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 16. | 5.5.12.6 | 81-82 | The information in this section was deleted in error from the October 19, 2015, version of the protocol. The information is being included in the July 25, 2017, version of the protocol to bring it back in line with the guidance in the Investigator Brochure regarding stopping olaparib 3 days prior to a planned surgery. The medical rationale for stopping olaparib 3 days prior to a planned surgery is purely a precautionary measure. Three days was chosen based on the half-life of olaparib which assumes that in 3 days most of the drug will have been eliminated. There are no data to suggest that olaparib has an impact on wound healing and no complications been reported perioperatively related to olaparib. |
| 17. | 6.4.7 | 96 | The risks below were added to the list of adverse events associated with olaparib based on the updated olaparib IB Edition 14 dated 10 March 2017. Immune System Disorders – Allergic reaction Skin and Subcutaneous Tissue Disorders – Dermatitis; Rash maculo-papular Bloating, which was added to the consent form in Amendment #3, was added to the list of Gastrointestinal Disorders. |
| 18. | 6.4.8 | 97 | Text was revised to match current CTEP template text for expedited reporting of adverse events. |
| 19. | 6.4.8.1 | 97 | Bullet 1: Text was revised to match current CTEP template text for expedited reporting methods. Bullet 4: An explanation about the review of CTEP-AERS reports by NRG Oncology and the NCI was added. Bullet 1: The instructions for submission of supporting documentation were clarified. |
| 20. | Table 8 | 99 | <ul> <li>The sponsor of the trial was changed from NCI to NRG Oncology because NRG Oncology is the sponsor for NSABP B-55/6-13.</li> <li>The table was revised to clarify that reports should be reported and submitted to the NCI and NRG Oncology.</li> </ul> |
| 21. | 6.4.9 | 100 | <ul> <li>Bullet 2 under reporting routine adverse events was revised to clarify that all ≥ grade 1 adverse events must be reported on the B-55/6-13 adverse event reporting form.</li> <li>Bullet 3 was added to remind sites that all adverse events reported via CTEP-AERS must also be reported on the B-55/6-13 adverse event forms in Medidata Rave.</li> </ul> |
| 22. | 6.4.10 | 105 | Paragraph 1: Text added to clarify that all SAEs are reported via CTEP-AERS and Medidata Rave. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 23. | 6.8 | 115 | Paragraph 2: |
| | | | <ul> <li>Text was added to clarify that pharmacokinetic<br/>sampling is being done only in patients<br/>participating in the pharmacokinetic component of<br/>the study.</li> </ul> |
| | | | • Bullets 3 and 5 were revised to clarify the time windows for each PK sampling collection. |
| 24. | 13.1 | 148 | Row 2: The Global Safety Physician's name and contact information was updated. |
| 25. | Appendices A, C, and D | 158-<br>200 | <ul> <li>Appendices were revised to match AstraZeneca's<br/>new Clinical Study Protocol template.</li> </ul> |
| | | | Appendix A Signatures was removed and subsequent appendices were relettered. References to appendices were revised throughout the protocol. |
| | | | Appendix D (Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law) was revised in line with the new AstraZeneca Clinical Study Protocol template: |
| | | | <ul> <li>Title was revised to "Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law."</li> <li>Table of contents was removed.</li> <li>The following sentence was added to the Introduction: "This Appendix describes the process to be followed in order to identify and appropriately report cases of Hy's Law. It is not intended to be a comprehensive guide to the management of elevated liver biochemistries."</li> <li>Definitions were revised.</li> </ul> |
| | | | <ul> <li>Section 6 "ACTIONS REQUIRED WHEN POTENTIAL HY'S LAW CRITERIA ARE MET BEFORE AND AFTER STARTING STUDY TREATMENT (NOT APPLICABLE)" was removed.</li> </ul> |

For Protocol Amendment #3 to: NSABP B-55/BIG 6-13

NCI Protocol #: NSABP B-55

Local Protocol #: NSABP B-55/BIG 6-13

NCI Version Date: 04/05/17

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | NSABP<br>PROTOCOL<br>B-55/BIG 6-13 | 1 | Amendment 3 was added to the Document History table with a NCI Version Date of April 05, 2017. |
| 2. | AstraZeneca<br>Clinical Study<br>Protocol | 2 | Amendment #3 was added to the AstraZeneca Clinical Study Protocol page. |
| 3. | Cancer Trials Support Unit (CTSU) Address and Contact Information | 21 | Column 1, Rows 1 and 2: Text updated to match CTSU template text regarding the requirement for submission of regulatory documentation through the CTSU portal. |
| 4. | 6.4.7 | 92 | The list of common adverse events associated with olaparib was revised based on changes requested in the Request for Rapid Amendment for olaparib dated March 10, 2017. • Weight loss was deleted from Investigations |

For Protocol Amendment #2 to: NSABP B-55/BIG 6-13

NCI Protocol #: NSABP B-55

Local Protocol #: NSABP B-55/BIG 6-13

NCI Version Date: 10/19/15

The following changes have been made from the July 22, 2014, version to the October 19, 2015, version of the protocol.

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | Section | T agv(s) | <ul> <li>The following changes have been made throughout the revised protocol:</li> <li>Investigational product changed to Study Treatment because this a double-blind study.</li> <li>Biobank changed to bio-repository.</li> <li>Twice daily added to clarify the dosing schedule for olaparib/placebo.</li> <li>Mammogram and breast MRI changed to mammogram and/or breast MRI to accommodate institutions that perform only one imaging technique.</li> <li>References to the FACIT-Fatigue and EORTC QLQ-C30 scale were changed to FACIT-Fatigue and EORTC QLQ-C30 questionnaire.</li> <li>Grammatical changes were made throughout the protocol.</li> </ul> |
| 2. | NSABP B-55 | 1 | <ul> <li>Not all changes are detailed in the Summary of Changes.</li> <li>NRG Oncology was added to the list of NCTN participating organizations.</li> <li>ECOG-ACRIN Medical Research Foundation, Inc. revised to ECOG-ACRIN Cancer Research Group.</li> <li>Address for NRG Oncology updated.</li> <li>Amendment #2 was added to the Document History table.</li> <li>NCI Version Date was changed from 07-22-14 to 10-19-15.</li> </ul> |
| 3. | AstraZeneca<br>Clinical Study<br>Protocol | 2 | The AstraZeneca Clinical Study Protocol page was updated with information from the Rest of World (RoW) protocol. |
| 4. | List of<br>Olympia<br>Protocol<br>Authors | 3-4 | A list of protocol authors of the B-55 (OlympiA) trial was added. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 5. | Study centre(s)<br>and number of<br>patients<br>planned | 5 | <ul> <li>The number of centres participating in the US and the rest of the world countries was changed from 300 to 500, and the study sample size was increased from 1320 to 1500 patients.</li> <li>Optional pharmacokinetic testing (RoW only) was added.</li> </ul> |
| 6. | Secondary<br>Objectives | 6 | <ul> <li>New primary cancers were added to Secondary Objective #3.</li> <li>A Secondary Objective (#6) was added for the pharmacokinetics study.</li> </ul> |
| 8. | Study delivery model | 7-8 | This new section describes who is sponsoring the trial in the U.S. and the RoW and how data will be collected. |
| 9. | Study design | 9 | <ul> <li>Paragraph 2: Hormone receptor status was added as a stratification factor.</li> <li>Paragraph 3: The description of treatment modality was clarified. Because this section is intended to be a summary of the study design, the description of adequate breast surgery was deleted and is found in Section 4.1 of the protocol.</li> <li>In Paragraph 2, the safety assessment "every 4 weeks for the following 5 months" was clarified as "up to week 24." Because this section is intended to be a summary of the study design, the description of follow-up testing and assessments was deleted. The information can be found in Section 3.1.</li> </ul> |
| 10. | Target patient population | 10 | Paragraph 1: Revised to include definition of ER and/or PgR HER2 negative patients. Patient populations categorized by adjuvant and neoadjuvant chemotherapy and TNBC and ER and/or PgR positive HER2 negative. |
| 11. | Hormone Receptor Positive/ HER2 negative Breast Cancer | 11 | Paragraph in the 07/22/14 version of the protocol describing inclusion of ER/PgR positive patients in the future has been deleted because ER and PgR positive patients are now eligible. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 12. | Germline BRCA1 and BRCA2 (gBRCA) testing | 11 | Section added to describe germline BRCA1 and BRCA2 testing requirements. |
| 13. | Central tumour analyses | 11 | New section added to describe central tumour analyses that will be done. The results of the central tumour analyses will be used for exploratory purposes in the context of the trial. |
| 14. | Study<br>treatment,<br>dosage and<br>mode of<br>administration | 11 | <ul> <li>Paragraph 2 deleted from revised protocol. Details included in Section 5.5.2.1.</li> <li>Comparator dosage and mode of administration section deleted from revised protocol. Information found in Section 5.5.3.</li> <li>Duration of treatment header deleted. Treatment regimen clarified.</li> </ul> |
| 15. | Stratification | 12 | <ul> <li>Paragraph 1, bullet 1: New stratification factor added to include hormone receptor positive patients.</li> <li>Paragraph 2: Statement added to clarify when unblinding will be allowed.</li> </ul> |
| 16. | Outcome(s) | 12 | <ul> <li>The word "variables" was deleted from the section heading and the bullet headings.</li> <li>Secondary Outcomes, hash mark 1: New primary cancers added.</li> <li>Secondary Outcomes, hash mark 2: All QOL instruments and scales being measured were added.</li> <li>Secondary Outcomes, hash mark 4: Pharmacokinetic analysis added as a secondary outcome.</li> <li>Safety outcomes: Electrocardiograms are no longer required after baseline so will not be followed as a safety outcome.</li> </ul> |
| 17. | Statistical methods | 13-15 | Sample size was revised and primary analysis information was added. The Statistical Methods section was shortened to include only an overview of the analyses to be done for the study. The complete description can be found in Section 12 of the protocol. |
| 18. | Pharmacoki-<br>netic analysis | 15 | New section added summarizing analysis of pharmacokinetic data. |
| 19. | Information<br>Resources | 23 | <ul> <li>Row 2, column 2: NRG Oncology mailing address updated.</li> <li>Row 6, column 3: CCD e-mail address revised to NRG Oncology e-mail address.</li> <li>Row 7, column 3: Reference to Patient Entry Guidelines located in Coordinator Online was deleted. Patient Entry information is found on the CTSU Information page.</li> <li>Row 9, columns 2 and 3: NSABP Division of Pathology updated to NRG Oncology Biospecimen Bank-Pittsburgh. E-mail address revised to NRG Oncology e-mail address.</li> <li>Row 2, column 3: SAE Reporting e-mail address revised to NRG Oncology e-mail address.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 20. | Cancer Trials<br>Support Unit | 25 | Row 2: CTSU phone number updated. Row 4: CCD e-mail address revised to NRG Oncology e-mail address. |
| 21. | List of<br>abbreviations<br>and definition<br>of terms | 26-30 | Abbreviations Added: CR Complete Response CRO Clinical Research Organization Hgb Hemoglobin Study treatment Study treatment is the treatment to which patient was randomized. In this study it is either olaparib or placebo |
| | | | Abbreviations Changed: CPS&EG Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS) - a disease scoring system EORTC QLQ-C30 The European Organisation for Research and Treatment of Cancer – Quality of Life Questionnaire – Core questions 30 |
| | | | Abbreviations Deleted: HRP high risk ER and/or PgR positive deleted because the abbreviation is not being used to describe this patient population in the protocol. IP Investigational Product LH Leutenising hormone PR Progesterone receptor SPAM (Study Procedures and Administration Manual) was deleted because the information found in the Study Procedures and Administration Manual is now found in the Laboratory Manual for RoW. |
| 22. | 1.1.1 | 31 | The Aaronson et al 1993 reference that was inadvertently added in the July 22, 2014, version of the protocol was deleted. |
| 23. | 1.1.2 | 32 | Hudis et al 2011 reference replaced with the correct reference of Dent et al 2007. |
| 24. | 1.1.5 | 33-34 | <ul> <li>New section added to provide rationale for including patients with ER and/or PgR HER2 negative breast cancer. Subsequent protocol sections renumbered.</li> <li>Description of olaparib and mechanism of action moved to Section 1.1.6.</li> </ul> |
| 25. | 1.1.6 | 34 | Information was part of Section 1.1.5 in the 07/22/14 version of the protocol and was moved to Section 1.1.6 of the revised protocol. Subsequent sections were renumbered. |
| 26. | 1.1.9 | 35 | Summary of clinical experience with olaparib deleted from the revised protocol. Current information can be found in the olaparib IB. |
| 27. | 1.1.9.1 | 36 | Study D0810C00020: The number of previous lines of chemotherapy patients received was clarified to indicate "3 or more" instead of "more than 3". |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 28. | 1.3 | 37 | • Paragraph 2, bullet 6: Second primary non-breast invasive malignancies defined. |
| | | 38 | • Paragraphs 1, 2, and 3: Information to support the inclusion of ER and/or PgR positive patients in the study and use of hormonal therapy was added. |
| | | | • Paragraph 4: Reason for following new cancers and overall survival for a minimum of 10 years was added. |
| 29. | 1.4 | 38-39 | • Paragraphs 1 and 2: The number of patients who have received olaparib across the olaparib development program was updated. |
| | | 39-40 | <ul> <li>Myelodysplastic syndrome/acute myeloid leukemia:<br/>Information on the number of cases of myelodysplastic<br/>syndrome/acute myeloid leukemia was updated.</li> </ul> |
| | | 41 | • Pneumonitis, paragraph 1: The number and details of cases of pneumonitis were updated. |
| | | 42-43 | • New malignancies other than MDS/AML: Information updated based on the olaparib IB dated 06-29-15. |
| 30. | 2.2 | 44 | <ul> <li>New primary cancers added to Secondary Objective #3.</li> <li>A Secondary Objective (#6) was added for the pharmacokinetics study.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 32. | 3.1 | 46-50<br>47<br>48-49 | <ul> <li>Section 3.1 was revised to delete the text describing the definitions for each of the patient populations eligible for the trial. The information is included in Section 4.1 Inclusion Criteria.</li> <li>Paragraph from 07/22/14 version of the protocol describing inclusion of ER/PgR positive patients in the future has been deleted because ER and PgR positive patients are now eligible.</li> <li>Details of germline BRCA1/2 mutation status, study treatment, stratification, and definition of adequate breast and axilla surgery from the 07/22/14 version of the protocol were deleted as they are found in other areas of the revised protocol.</li> <li>Paragraph 1: Clarification of when radiological examinations can be replaced by clinical examination and ultrasound. Assessment schedule to be followed if study treatment discontinued early was deleted. Information in other sections of protocol.</li> <li>Paragraph 2: Imaging requirement was clarified to include other imaging allowed in addition a CT/MRI scan. Definition of subsequent therapies was added.</li> <li>Paragraph 1: Second sentence was deleted because it was duplicative.</li> </ul> |
| | | 49-50 | <ul> <li>Instructions added for patient follow-up after premature<br/>discontinuation of treatment or if treatment is discontinued<br/>because an IDFS endpoint is met or discontinuation if an<br/>IDFS endpoint is not met.</li> </ul> |
| 33. | Study Flow<br>Chart | | <ul> <li>First box revised to clarify ICF is signed by patients with unknown BRCA status.</li> <li>Neoadjuvant chemotherapy, Surgery, and Adjuvant Chemotherapy text boxes revised to reflect key inclusion criteria.</li> <li>Description of eligible patient population added to the Non-Path CR text box following the Surgery text box.</li> <li>Informed consent for participation in the study (after surgery or adjuvant chemotherapy) was clarified to indicate that informed consent is obtained from patients with known gBRCA mutation status.</li> <li>Time period in which a patient should be randomized after last treatment was revised.</li> <li>Time point for next mammogram and/or breast MRI changed from randomization to day 1.</li> <li>Clarification of when study will end was added.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 34. | Table 1 | 53 | <ul> <li>Row 1, column 2 header changed to clarify that the patient can sign the informed consent form prior, during, or after neoadjuvant or adjuvant chemotherapy or radiotherapy.</li> <li>Row 1, column 3 header changed to clarify screening requirements are for patients with confirmed BRCA status by Myriad, or if known, prior to study entry (done by local testing).</li> <li>Row 3, column 1: Date of birth added as information collected as part of demographics.</li> <li>Row 6, column 2: Second asterisk added.</li> <li>Rows 19 and 20, column 1: The archival tumour was clarified to indicate it is to be FFPE.</li> <li>Row 20, Column 1: Footnote l deleted. Subsequent footnotes relettered.</li> </ul> |
| | | 54 | <ul> <li>Row 3, Columns 1-3: Collection of "Family history of cancer" added. The exact distribution of de novo germline BRCA mutations versus inherited germline BRCA mutations in the studied target populations with HER2 negative breast cancer and a confirmed germline mutation in BRCA1 or BRCA2 remains unknown. Knowledge of these proportions in the target breast cancer population studies might inform and refine future recommendations for tailoring genetic testing in such patients.</li> <li>Footnote a revised to clarify the Part 1 time period for patients that require Myriad gBRCA testing.</li> <li>Footnote b revised to clarify recommendation for when to consent patients that require Myriad gBRCA testing.</li> <li>Footnote d revised to add components of CPS&amp;EG score that are to be collected.</li> <li>Footnote g revised to indicate ECG assessment is to be done within 28 days before randomization.</li> <li>Footnote h: Clarified to indicate that dipstick is required.</li> <li>Footnote i: Women who must have a pregnancy test done was clarified. The timing for pregnancy testing was revised from 28 days prior to starting treatment to 28 days prior to randomization for consistency throughout the protocol.</li> <li>Footnote j was revised to clarify that patients with a known BRCA status should be consented within 28 days prior to randomisation.</li> <li>Footnote k was revised clarify the tumour sample</li> </ul> |
| | | 55 | <ul> <li>submission requirements for participation in the study.</li> <li>Footnote I, "Neoadjuvant patients only," was deleted from the 07/22/14 version of the protocol. Subsequent footnotes were relettered.</li> <li>New footnote I: Description of patients considered at high risk of having disseminated disease was revised. Timing of will mammogram and/or breast MRI added.</li> <li>Footnote o was added to clarify that coagulation analysis is only required at baseline.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 35. | Table 2 | 56 | • Row 4, columns 7 and 8: Visit window changed from ±2 weeks to +2 weeks. |
| | | 57 | <ul> <li>"ECG as clinically indicated" deleted from Table 2. ECG only required prior to randomisation.</li> <li>New Rows 12-14 added for collection of blood samples for</li> </ul> |
| | | | pharmacokinetic analysis and biomarker and tumour samples at recurrence. |
| | | | • Footnote a: The timing for pregnancy testing was revised to clarify that a pregnancy test must be performed prior to the first dose of study treatment on Day 1. |
| | | | <ul> <li>Footnote c revised to clarify when safety blood samples<br/>have to be repeated, and coagulation analysis requirement<br/>deleted.</li> </ul> |
| | | | • Footnote e: Clarification of when breast imaging to be performed. |
| | | | <ul> <li>Footnote f deleted: Timing of QOL assessments on table.</li> <li>Subsequent footnotes relettered.</li> </ul> |
| | | | • Footnote g: Follow-up requirements when study treatment discontinued early added. Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse. |
| | | | <ul> <li>Footnote h was added to describe the blood collection time points for the pharmacokinetic samples.</li> <li>Footnote i: Time point for collection of biomarker analysis samples added.</li> </ul> |
| | | 59 | • Footnote k added to give information about the optional tumour biopsy at recurrence. |
| | | | • The Note after the footnotes was deleted. Revised information included in footnote g. |
| 36. | Table 3 | 60 | <ul> <li>The Visit Number and Month schedules were expanded to clarify the assessment time points. The Visit Window columns were revised.</li> <li>A new Row 13, SAE, was added.</li> </ul> |
| | | 61 | • Footnote a: Clarification of when breast imaging to be performed. |
| | | | <ul> <li>Footnote b: Subsequent therapies that are to be collected were clarified.</li> </ul> |
| | | | • Footnote c deleted because timing of QOL assessments on table. Subsequent footnotes relettered. |
| | | | Footnote e: Instructions for SAE reporting after completion of study treatment added. |
| 37. | 3.2.1 | 62 | ER and/PgR HER2 negative patients added to study design because these patients are eligible. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 38. | 3.2.3 | 63 64-65 | <ul> <li>Paragraph 1, sample size changed to 1500.</li> <li>Bullet 1: BRCA mutation clarified to indicate germline BRCA mutations.</li> <li>Hash marks 1 and 2: Central laboratory deleted as descriptor of Myriad.</li> <li>Bullet 1: Phenotypic tumour selection revised to indicate that TNBC and ER and/or PgR positive HER2 negative are eligible.</li> <li>Bullet 1, paragraph 2 from July 22, 2014, version of the protocol was deleted because ER and/or PgR HER2 patients are able to participate.</li> <li>Bullet 2, #1 and #2: Definitions of high risk of recurrence for patients based on treatment was revised.</li> </ul> |
| 39. | 4. | 66 | A second asterisk was added to paragraph 3. |
| 40. | 4.1 | 66<br>66-67<br>67<br>68<br>69 | <ul> <li>A second asterisk was added to criteria 1-2, 4, 11b, and 12.</li> <li>Criteria 3 and 4 revised to include ER and/or PgR positive, HER2 negative patients. HER2 negative requirements revised to match ASCO/CAP definition in criterion 4, and text added to clarify patient eligibility of patients with multifocal or multicentric or synchronous bilateral invasive disease. Subsequent criteria renumbered.</li> <li>A new criterion 3 was added to clarify nodal status required for patients who received neoadjuvant or adjuvant chemotherapy. Subsequent criteria renumbered.</li> <li>Criterion 5 revised to clarify the BRCA mutation is germline and which gBRCA testing and results can be used for determining eligibility.</li> <li>Criterion 6 revised to define adequate breast surgery and definition of axilla surgery.</li> <li>Criterion 7: Instruction added that all neoadjuvant chemotherapy must be given prior to surgery.</li> <li>Criterion 8 revised to clarify when blood transfusions can occur and that patients with elevated ALT/AST or ALP require additional testing to rule out metastatic breast cancer.</li> <li>Criterion 9: Plasma added as sample that can be used for creatinine testing.</li> <li>Criterion 11a revised to to state that a negative urine or serum pregnancy test must be done within 28 days prior to randomization instead of 7. Criterion 11b was added in response to a request from the FDA to include contraception use as an inclusion criterion.</li> </ul> |
| | | 71 | <ul> <li>Criterion 13 revised to clarify tumour sample requirements.</li> <li>Criterion 14 added to indicate timeframe within which patients must be randomised.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 41. | 4.2 | 71<br>71-72<br>72 | <ul> <li>A second asterisk was added to criteria 1, 3-7, 13, and 16, 18-20.</li> <li>Criterion 2: Definition of <i>BRCA</i> mutation status clarified.</li> <li>Criterion 4 was revised to clarify definition of patients considered at high risk of having disseminated disease. Imaging requirements to rule out metastatic breast cancer clarified.</li> <li>Criterion 7: Second primary malignancy exceptions clarified.</li> <li>Criteria 9, 10, and 14 were revised to clarify when procedures should be done, i.e., prior to randomisation and not prior to starting study treatment.</li> <li>Criterion 11: Instruction added that there is a minimum washout period prior to starting olaparib when using CYP3A4 inhibitors. Specific information can be found in Appendix I.</li> <li>Criterion 13: Exclusion criterion for MDS/AML clarified.</li> </ul> |
| 42. | 5.1.1 | 73 | Contraception requirements for female and male patients revised based on the olaparib IB dated 06-29-15. |
| 43. | 5.2 | 73-74 | Numbers 1-7: Patient enrolment, randomisation, and initiation of study treatment instructions clarified. |
| 44. | 5.2.4 | 76<br>77 | <ul> <li>Paragraph 1: Text added as to when randomization can take place.</li> <li>Paragraph 2: Hormone receptor status added as a stratification factor.</li> <li>Paragraph 1: Patients may start study therapy up to 21 days from randomization.</li> <li>Paragraph 2 revised to clarify that when incorrect information entered at randomisation, the correct information should be recorded in the eCRF not the clinical database.</li> </ul> |
| 45. | 5.4.2 | 78-79 | Examples of situations for unblinding and not unblinding study treatment added. |
| 46. | 5.5.2.1<br>(Section<br>5.5.7.1 in<br>07/22/14<br>version) | 80 | <ul> <li>B-55/6-13 olaparib doses presented in table format (see Table 5).</li> <li>Paragraph 1 revised to include instruction that patients should not take two doses at the same time.</li> </ul> |
| 47. | 5.5.3 | 81 | <ul> <li>Paragraph 3 under How Supplied: Drug kit contents clarified by CTEP Pharmaceuticals Management Branch (PMB).</li> <li>Stability: Stability of study treatment updated by PMB.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 48. | 5.5.4 | 83 | Instructions for obtaining an olaparib IB from CTSU added. |
| 49. | 5.5.5 | 83 | Procurement of olaparib instructions updated by PMB. |
| 50. | 5.5.6<br>(Section 5.5.8<br>in 07/22/14<br>version) | 84 | Section moved and paragraph 2 added by the PMB. |
| 51. | 5.5.8 | 84-85 | Return of olaparib/placebo instructions updated by PMB. |
| 52. | 5.5.9 | 86 | <ul> <li>Bullets 4 and 13: Patient ID number example changed to match B-55/6-15 Patient ID format.</li> <li>Bullet 8: Instruction added to discard bottle contents after 90 days of opening.</li> <li>Paragraph 1: Information from bottle label that is to be recorded on Oral DARF was added by PMB.</li> </ul> |
| 53. | 5.5.10 | 87 | General instructions for managing toxicity were added. |
| 54. | 5.5.10.1 | 87 | Instructions for discontinuing study therapy following breast cancer recurrence or second primary cancer. |
| 55. | 5.5.10.2 | 87<br>88 | <ul> <li>Clarification of dose reduction and re-escalation process.</li> <li>Table 6 showing olaparib/placebo dose levels added.</li> <li>Information in the "Management of toxicity" section of the 07/22/14 version of the protocol was combined into Table 7 of the revised protocol.</li> </ul> |
| 56. | 5.5.10.3 | 90 89-92 | <ul> <li>Table 5 from 07/22/14 version of the protocol deleted. Subsequent tables were renumbered. Instructions on managing hematological toxicities are found on Table 7.</li> <li>Information from the Management of haematological toxicity section in the 07/22/14 of the protocol was added to the Hematologic Toxicity section of Table 7.</li> </ul> |
| 57. | 5.5.10.5<br>(Section<br>5.5.10.1 in<br>07/22/14<br>version) | 93 | Paragraph 1 from 07/22/14 version of the protocol describing frequency of nausea and vomiting deleted as this section is intended to address management of the toxicities. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 58. | 5.6 | 93 | <ul> <li>Paragraph 1: Instructions clarified as to when concomitant medications can be given.</li> <li>Paragraph 2 added to specify that bisphosphonates or denosumab are allowed during study treatment and follow-up.</li> <li>Paragraph 2: Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse.</li> <li>Paragraph 3: Prohibited medications during study treatment and follow-up were added.</li> <li>Paragraph 4: Instructions regarding initiation of subsequent anti-cancer treatment after breast cancer recurrence and the information to be collected were added.</li> </ul> |
| 59. | 5.6.1 | 94 | Section on administration of endocrine therapy added. Subsequent sections renumbered. |
| 60. | 5.6.2 | 94-95 | The summary of olaparib and CYP3A4 interaction was updated. |
| 61. | 5.6.3 | 95 | Information on effect of olaparib on other drugs added. |
| 62. | 5.6.4 | 96 | Section 5.6.4 from the 07/22/14 version of the protocol was deleted. Information addressed in Section 5.6. Replaced with Interaction of olaparib and specific co-medications. |
| 63. | 5.6.6 | 96 | Use of other oral anticoagulants besides subcutaneous heparin is allowed. |
| 64. | 5.6.7 | 96 | Protocol section added to clarify the use of live virus and bacterial vaccines while taking study treatment. |
| 65. | 5.7 | 96 | <ul> <li>Paragraph 1: The time period of study treatment was added.</li> <li>Paragraph 2: Instructions for tablet counts were changed from will to should.</li> </ul> |
| 66. | 5.7.1 | 97 | Accountability instructions updated by the PMB. |
| 67. | 5.8 | 97 | Bullets 4 and 10 were added as reasons for which a patient may be discontinued from study treatment |
| 68. | 5.8.1 | 98-99 | Section revised to provide instructions for patient follow-up after discontinuation of study treatment and information to be collected. |
| 69. | 6.1.2 | 101 | Information about Expected/Delinquency Report deleted because report no longer available on Coordinator Online. |

| | Section | Page(s) | Change |
|---|---|---|---|
| 70. | 6.2.1 | 102 | <ul> <li>Paragraph 1, revised to clarify when procedures should be done, i.e., prior to randomization and not prior to first dose of study treatment.</li> <li>New bullet 7: Family history of cancer to be collected.</li> </ul> |
| | | | • Bullet 10 revised to state that an ECG should be done within |
| | | | 28 days prior to randomisation and not 7 days prior to start of study treatment. |
| | | | • New bullet 13: Instructions for performing breast imaging added. |
| | | | • Bullet 14 revised to clarify that pregnancy testing is required within 28 days prior to randomisation and on Day 1 before starting study treatment. |
| | | | <ul> <li>Bullet 15 revised to add location of instructions for<br/>calculating the CPS&amp;EG score.</li> </ul> |
| | | 103 | • Bullet 1: Additional information added to describe germline <i>BRCA1/2</i> mutation status determination. |
| | | 104 | • Bullet 1: Change made to clarify that only serious adverse events must be collected from time of consent. |
| 71. | 6.2.2 | 104 | • Bullet 1: Instruction for reporting findings of physical exam clarified. |
| | | | • Bullets 2 and 3: Timing of assessments clarified. |
| | | | • Bullet from 07/22/14 version of protocol for ECG any time if clinically indicated was deleted because this is no longer a requirement. |
| | | 105 | • Bullet 1 revised to clarify when safety blood samples should be collected. |
| | | | • Bullet for coagulation deleted because coagulation assessments are not required during study treatment. |
| | | | • Bullets 1, 3, and 6: Timing of assessments clarified. |
| | | | • Bullet 2: Added to indicate race and ethnicity of patients is collected. |
| | | | • Bullet 5 added for collection of optional pharmacokinetic samples. |
| | | | • Bullet 7 added for pharmacokinetic samples being collected in RoW patients. |
| | | | Bullet 10: Clarification of when breast imaging to be performed. |
| | | | <ul> <li>Bullet 11 revised to indicate that return of unused study<br/>treatment is required.</li> </ul> |
| 72. | 6.2.3 | 105-<br>106 | Paragraphs 1-4: Assessment schedules and data to be collected are clarified. |
| 73. | 6.2.4 | 106 | Details of long term safety collection were added to Section 6.4.9. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 74. | 6.2.5 | 106-<br>107 | <ul> <li>Paragraph 1: Data cut off for primary analysis will occur after a minimum of 330 IDFS events or last randomised patient has been followed for a minimum of 24 months, whichever occurs latest.</li> <li>Paragraph 1: Sentence with duplicative instructions was</li> </ul> |
| 7.5 | 6.2.1 | | deleted. |
| 75. | 6.3.1 | 107<br>107-<br>108 | <ul> <li>Paragraph 2: Mammograms and/or breast MRIs are to continue for approximately 10 years beginning 6 months after day 1.</li> <li>Protocol revised to explain the assessment schedules to be followed if a patient has a recurrence. Data to be collected is also described.</li> </ul> |
| 76. | 6.4.6 | 109 | Study phase clarified in paragraph 1. |
| 77. | 6.4.7 | 110 | The list of adverse events associated with olaparib was revised to match the risks provided by CTEP in the Request for Rapid Amendment dated April 7, 2015. The CAEPR list was not included as NRG Oncology is the IND holder for the trial. The risks of "edema limbs" and "cough" were added to the expected risks for olaparib. |
| 78. | 6.4.9 | 113<br>115<br>116 | <ul> <li>Paragraph 1 revised to clarify timing of reporting serious adverse events.</li> <li>Paragraph 2: Instructions added for reporting MDA/AML or new primary malignancy.</li> <li>Paragraph 3: Revised to be consistent with Section 6.2.1.</li> <li>Paragraph 7: Protocol revised to clarify that AEs must be collected and recorded in the eCRF and then submitted.</li> <li>Paragraphs 1 and 3: Protocol revised to clarify that AEs must be collected and recorded in the eCRF and then submitted.</li> <li>Disease recurrence: First sentence deleted. Not applicable to an adjuvant trial.</li> <li>Lack of efficacy: Section deleted from the 07/22/14 version of the protocol. Not applicable to an adjuvant trial.</li> <li>Deaths, bullets 1 and 2: Disease recurrence or progression changed to disease under study recurrence or progression to indicate recurrence or progression related to breast cancer.</li> </ul> |
| 79. | 6.4.12 | 120 | The list of assessments to be done in a physical examination was deleted to allow the investigator to perform a physical examination based on local standards. |
| 80. | 6.4.13.1 | 120 | Paragraph 1 revised to clarify that an ECG is required 28 days prior to randomisation. ECG no longer required to be done after baseline testing. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 81. | 6.4.14.1 | 121 | The requirement to rest 10 minutes on a bed before taking blood pressure and pulse was deleted. |
| 82. | 6.4.15.1 | 121 | The timing for pregnancy testing was revised from within 7 days prior to start of study treatment to within 28 days prior to randomization for consistency throughout the protocol. Instruction added that results must be available before study treatment started. |
| 83. | 6.5.1 | 122 | Last sentence deleted. Information in Section 3.2.2. |
| 84. | 6.5.2 | 122 | EORTC QLQ-C30 subscales clarified. |
| 85. | 6.5.3 | 122-<br>123 | Paragraph 2: Protocol changed to specify that a trained person must administer the PRO questionnaires and not a specific individual. |
| | | 123 | • Paragraph 1, bullet 1: PRO questionnaires are to be completed at the clinical visit. |
| 86. | 6.6.1<br>Table 9 | 124 | <ul> <li>Text added under "Archival tumour sample" to clarify what archival tumour samples are required for participation on the study. Footnote for mandatory tumour sample requirements was revised to clarify the tumour sample submission requirements for neoadjuvant and adjuvant patients.</li> <li>Blood samples for biomarker analysis visit changed to Day 1 prior to first dose of study treatment instead of randomisation to match Table 2.</li> </ul> |
| 87. | 6.6.2 | 125 | <ul> <li>Paragraph 1: Information on the number of samples to be collected and use of each one was added.</li> <li>Paragraph 2: Text revised to clarify how <i>BRCA</i> results are to be entered in the database.</li> </ul> |
| 88. | 6.6.2.1 | 126 | Text from Section 6.6.2.1 of the 07/22/14 version of the protocol deleted because information covered in Section 6.6.2. Subsequent sections renumbered. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| | | - | |
| 94. | 6.8 | 129-<br>130 | The following new sections were added to the revised protocol. Subsequent section was renumbered. 6.8 Pharmacokinetics (optional) 6.8.1 Pharmacokinetic samples 6.8.2 Collection of samples 6.8.3 Determination of drug concentration |
| 95. | 7.1 | 130 | The maximum volume of blood that can be drawn from each patient was changed from 198 mL to 208 mL to include the subset of patients having pharmacokinetic samples collected. |
| 96. | 7.1<br>Table 10 | 131 | <ul> <li>Collection time points for biomarkers changed to be day 1 instead of randomisation. Samples are to be drawn at 30 days post study treatment discontinuation.</li> <li>Pharmacokinetic sample added to table to include sample volume, number of samples, and total sample volume.</li> </ul> |
| 97. | 7.2.2 | 132 | Information about the use, analysis, and destruction of the pharmacokinetic samples added. |
| 98. | 7.5 | 133 | <ul> <li>Paragraph 4 revised to describe the mandatory tumour sample requirements of tumour sample submission for neoadjuvant and adjuvant patients.</li> <li>Paragraph 1: If a patient withdraws use of tumour sample collected at the time of relapse, the patient can continue in the study.</li> <li>Paragraph 2: If a patient withdraws use of pharmacokinetics samples, the patient can continue in the study.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 99. | 8.3 | 135 | Paragraph 7: BIG/Partners added to AstraZeneca as groups responsible for submission of safety updates/reports to regulatory authorities. |
| 100. | 9.3 | 138 | Bullet 1: Monitoring of study includes verification that appropriate version of consent form used and was signed and dated prior to any study procedures. |
| 101. | 9.3.1 | 138 | Section deleted to eliminate confusion at sites because information not applicable to conduct of study in US. |
| 102. | 9.4 | 138 | Section deleted to eliminate confusion at sites because information not applicable to conduct of study in US. Subsequent section renumbered. |
| 103. | 9.4.1 | 138 | Section deleted to eliminate confusion at sites because information not applicable to conduct of study in US. |
| 104. | 9.4<br>(Section 9.5 in 07/22/14 version) | 138 | Paragraph 3 added to describe that end of study will occur 10 years following the randomisation of the last patient, and patients will be followed until 10 years after the randomisation of the last patient. |
| 105. | 10. | 139 | <ul> <li>Paragraph 2: Frontier Science added as the party who will reconcile B-55/6-13 data.</li> <li>Paragraph 3: Change made to clarify that Frontier Science and not AstraZeneca will be responsible for coding.</li> <li>Paragraph 4: Sentence added to clarify that data management procedures are found in the Data Management Plan for the study.</li> <li>Paragraph 6: Statement added that the roles and responsibilities of staff involved in the data management process can be found in the Data Management Plan.</li> <li>Text from the 07/22/14 version of the protocol about data management relative to the B-55/6-13 genetic research was deleted. It is covered in the Clinical Study Report.</li> </ul> |
| 106. | 11.1.1 | 140 | <ul> <li>Bullet 6: Examples and exceptions to second primary non-breast invasive malignancies added.</li> <li>Paragraph 3: Local recurrence events are to be based on an objective finding. Not all investigators consider the tests and procedures listed as clinical assessments.</li> <li>Paragraph 4: Imaging examination can also be used to determine distant recurrence</li> <li>Paragraph 1: The date of the earliest objective finding will be used for the date of the new cancer for the analysis.</li> <li>Paragraph 5: Definition of disease evaluation clarified.</li> </ul> |
| 107. | 11.1.2.3 | 142-<br>143 | Paragraph 5: Definition of disease evaluation clarified. The cancers to be collected as part of data collection for the study expanded. Explanations of patient who will or will not be included in the data analysis were clarified. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 108. | 11.2 | 143 | ECG not included as safety variable because ECG only done at baseline. |
| 109. | 11.4 | 143 | The location where pharmacokinetic analysis will be done and the process for calculation or derivation of pharmacokinetic variables were added. |
| 110. | 12.1.1 | 144 | #2: Sample size for the mature cohort ITT population was revised from 660 to 750. |
| 111. | 12.1.2<br>Table 11 | 144-<br>145 | <ul> <li>New cancers added to list under Efficacy data – Final.</li> <li>Pharmacokinetics data added as an Outcome Variable.</li> </ul> |
| 112. | 12.1.3 | 145 | PK analysis set section was added. |
| 113. | 12.2.1.1 | 145-<br>149 | Changes to the methods for analysis of the study data were based on recommendations from the U.S. Food and Drug Administration. Section 12.2.1 was divided into 4 subsections in the revised protocol. |
| | | 145 | <ul> <li>Paragraph 1: Time point when primary analysis of IDFS<br/>will occur was described.</li> </ul> |
| | | 146 | <ul> <li>Paragraph 1: IDFS analyzed using a Cox proportional<br/>hazard model instead of the log-rank test.</li> </ul> |
| 114. | 12.2.1.2 | 146 | Paragraph 2: Description of how patients mis-stratified will be analyzed. |
| 115. | 12.2.1.3 | 147 | <ul> <li>The following have been added as subgroups of primary interest for analysis:</li> <li>Bullets 1 and 4: Hormone receptor status and BRCA mutation type added.</li> <li>Bullet 6: BRCA status by prior platinum therapy setting added.</li> <li>The following are additional subgroups to be analyzed (as known before start of study medication) or revised subgroups.</li> <li>Bullet 3: Bullet shortened to bilateral oophorectomy (Yes/No).</li> <li>Bullet 5: CPS+EG score groups revised.</li> <li>Bullet for BRCA mutation type from 07/22/14 version of the protocol deleted. Included in subgroup of primary interest.</li> <li>Bullet 6: The age groups that will be used in stratification were added to Age at randomisation.</li> <li>Bullet 8: Geographic region changed to Sponsor (AZ; NRG Oncology)</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 116. | 12.2.2 | 149<br>150 | <ul> <li>Paragraph 3: Primary analysis for IDFS clarified.</li> <li>Incidence of contralateral invasive breast or new ovarian cancer section heading revised to include additional cancers that will be included in study analyses.</li> <li>Paragraph 1: New cancers added to those that will be collected and analyzed.</li> <li>Paragraph 2: Patients who will be excluded from analysis is described.</li> <li>Paragraph 3: Analysis of cumulative incidence of new primary cancers compared between treatment groups is</li> </ul> |
| 117. | 12.2.3.1 | | described. Paragraph 1: Statement that analyses of Patient Reported Outcomes will be conducted on the ITT population added. |
| 118. | 12.2.3.2 | 152<br>153<br>153-<br>154 | <ul> <li>Paragraph 2: Additional covariate to be used in the analysis of the primary endpoint of fatigue was added.</li> <li>Sample size consideration revised based on addition of ER and/or PgR positive patients.</li> <li>Missing PRO data section revised to include how missing data will be analyzed based on whether or not a missing data mechanism is detected.</li> </ul> |
| 119. | 12.2.3.3 | 154 | A new section for Pharmacokinetic analysis was added. |
| 121. | 12.2.6 | 159 | Interim analysis information and Table 12 updated based on increase in sample size and inclusion of ER and/or PgR positive HER2 negative patients. |
| 122. | 12.2.7 | 159-<br>162<br>160<br>161 | <ul> <li>Sample size justification section was revised to update the sample size of the study, when primary analysis would be done, and the estimated time for accrual.</li> <li>Table 13 with the estimated accrual pattern for the study was added.</li> <li>Table 14 was added to provide the estimated annual hazard rates used in the calculation of the sample size.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 123. | 14. | 168- | References added: |
| | | 176 | Atchley et al 2008 |
| | | | Cortazar et al 2014 |
| | | | Dent et al 2007 |
| | | | Fine and Gray 1999 |
| | | | Gupta et al 2007 |
| | | | Honrado et al 2006 |
| | | | Morton et al 2013 |
| | | | Nardone et al 2015 |
| | | | Schiewer et al 2013 |
| | | | Swain et al 2013 |
| | | | Tryggvadottir et al 2013 |
| | | | Vay et al 2011 |
| | | | Zhang et al 2013 |
| | | | References deleted: |
| | | | Berry et al 1991 |
| | | | FDA Guidance for Industry 2012 |
| | | | Hudis et al 2011 |
| | | | Selke et al 1983 |
| | | | Reference corrected or updated: |
| | | | Celle D et al 2002 |
| | | | Ganz et al 1998A and Ganz et al 1998B |
| | | | Ganz et al 2011A and Ganz et al 2011B |
| | | | Kaufman et al 2014 |
| | | | Year of publication for Glimm et al and for Stone corrected |
| | | | from 2009 to 2010. |
| 124. | Appendix E | 201 | Bullets 2 and 3: AE/SAE reporting instructions revised for U.S. |
| | | | reporting process. |
| 125. | Appendix F | 204- | Paragraph 1: Revised to specify length of time birth control |
| | | 205 | that must be used for female and male patients. |
| | | | • Paragraph 2: Specific birth control information for male |
| | | | patients was added. |
| | | | Acceptable non-hormonal birth control methods were |
| | | | updated to provide clarification that true abstinence is |
| | | | expected in line with preferred and usual life style |
| | | | according to patient choice. The wording also provides |
| | | | clear guidance on contraception methods that cannot be |
| | | | classified as true abstinence. |
| | | | • Male condoms no longer need to be used with a spermicide. |
| | | | <ul> <li>Additional acceptable hormonal methods were added.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 126. | Appendix I | 215<br>216-<br>217 | <ul> <li>Potent inhibitors of CYP3A4 information updated.</li> <li>"Effect of olaparib on other drugs" and "Interaction of olaparib and specific co-medications" added.</li> </ul> |
| 127. | Appendix J | 218-<br>219 | A new appendix was added for instructions on calculation of the CPS & EG score. |
| 128. | Sample<br>Consent Forms | | Consent form changes are outlined in the Summary of Changes for each B-55/6-13 consent form. |

For Protocol Amendment #1 to: NSABP B-55/BIG 6-13

NCI Protocol #: NSABP B-55

Local Protocol #: NSABP B-55/BIG 6-13

NCI Version Date: July 22, 2014

Protocol Title: A Randomised, Double-Blind, Parallel Group, Placebo-Controlled Multi-Centre Phase III Study to Assess the Efficacy and Safety of Olaparib Versus Placebo as Adjuvant Treatment in Patients with Germline BRCA1/2 Mutations and High Risk HER2 Negative Primary Breast Cancer Who Have Completed Definitive Local Treatment and Neoadjuvant or Adjuvant Chemotherapy

The following changes have been made from the May 12, 2014, version to the July 22, 2014,

version of the protocol and informed consent documents.

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | 1. Global | | The following changes have been made throughout the revised protocol: |
| | | | <ul> <li>The NSABP and the NSABP Operations Center were changed<br/>to NRG Oncology, where appropriate.</li> </ul> |
| | | | • As part of the restructuring of the cooperative groups, the name of the NSABP Biostatistical Center has been changed to the NRG Oncology Statistics and Data Management Center (SDMC). All references to NSABP Biostatistical Center have been changed to NRG Oncology SDMC. |
| | | | <ul> <li>Divisions are now referred to as Departments within NRG Oncology. Division has been changed to Department where appropriate.</li> <li>QOL changed to QoL for consistency throughout the</li> </ul> |
| | | | protocol. |
| 2. | NSABP | 1 | • The ClinicalTrials.gov ID number for this trial was added. |
| | PROTOCOL B-<br>55/BIG 6-13<br>Title Page | | <ul> <li>The NCTN participating organizations descriptions were<br/>revised according to CTEP's standard language.</li> </ul> |
| | | | • The version date was changed from May 12, 2014, to July 22, 2014. |
| | | | <ul> <li>The IND sponsor was changed from the NSABP to NRG<br/>Oncology, Inc.</li> </ul> |
| | | | <ul> <li>A Document History table was added for consistency with<br/>other NRG Oncology protocols.</li> </ul> |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 3. | Information | 19 | The phone number for CTSU was updated. |
| | Resources | | • The website for the B-55/6-13 Pathology and Correlative Science Instructions was updated because the instructions are only found on the CTSU website. |
| | | | • Contact information for the NSABP Division of Pathology was added. |
| 4. | Information<br>Resources | 21 | The website for the location of data forms has been changed from NSABP to CTSU. |
| 5. | Cancer Trials Support Unit (CTSU) Address And Contact Information | 22 | The CTSU table was revised in Row 2, Columns 1 and 2 to include updated standard language from CTSU. |
| 6. | List Of Abbreviations And Definitions Of Terms | 24, 26 | CTEP-IAM: CTEP Identity and Access Management and NCTN:<br>National Clinical Trials Network were added to the list. |
| 7. | 1.4 | 34 | Aaronson et al reference that was inadvertently included in list of references was deleted. |
| 8. | 4.1<br>Criterion #8 | 57 | The instruction for patients with a screening ALT/AST or ALP above the institutional upper limit of normal was changed from "must" to "should" be consistent with instructions in footnote m of Table 1. |
| 9. | 5.2.1 and 5.2.2 | 58-59 | Sections 5.2.1 and 5.2.2 were revised to include updated text from CTSU for investigator and associate registration procedures. |
| 10. | 5.2.3 | 60-61 | <ul> <li>Site registration procedures were added and include the standard language provided by CTSU for obtaining IRB approval, downloading site registration documents, submitting regulatory documents, and checking site registration status.</li> <li>Subsequent sections were renumbered.</li> </ul> |
| 11. | 5.2.5 | 63 | Section revised to include updated standard language from CTSU regarding patient enrollment and OPEN. |
| 12. | 6.1.1 | 79 | Instructions were revised and the second bullet was deleted. |
| 13. | 6.4.1 | 85 | IND sponsor updated from the NSABP to NRG Oncology, Inc. |
| 14. | 6.4.7 | 86 | A new risk, mucositis oral, was added to the adverse events associated with olaparib as requested by AstraZeneca due to an updated olaparib IB. |

| # | Section | Page(s) | Change |
|---|---|---|---|
| 18. | 8.3 | 109 | CIRB was defined as this is the only instance of the use of CIRB in the protocol. |
| 19. | 13.1 | 134-<br>135 | <ul> <li>Contact information for was updated.</li> <li>Phone number for 24-hour emergency cover at NRG Oncology updated.</li> </ul> |
| 20. | 13.3.2 | 136 | The website where the Pregnancy Information Form is located was updated from NSABP to CTEP. |

#### NRG ONCOLOGY

# NSABP PROTOCOL B-55/BIG 6-13

ClinicalTrials.gov NCT02032823

A Randomised, Double-Blind, Parallel Group, Placebo-Controlled Multi-Centre Phase III Study to Assess the Efficacy and Safety of Olaparib Versus Placebo as Adjuvant Treatment in Patients with Germline BRCA1/2 Mutations and High Risk HER2 Negative Primary Breast Cancer Who Have Completed Definitive Local Treatment and Neoadjuvant or Adjuvant Chemotherapy

This trial is part of the National Clinical Trials Network (NCTN) program, which is sponsored by the National Cancer Institute (NCI). The trial will be led by NRG Oncology with the participation of the network of NCTN organizations (U.S. Institutions only): the Alliance for Clinical Trials in Oncology, ECOG-ACRIN Cancer Research Group, NRG Oncology, and SWOG.



NRG Oncology Statistics and **Data Management Center** 

### CLINICAL COORDINATING DEPARTMENT: Redacted

(For Clinical Questions Only)

### KEY STUDY PERSONNEL

NRG Oncology Group Chairman: NRG Oncology Breast Committee Chair:

Protocol Chairs:

Protocol Officer:

Behavioral and Health Outcomes Officer:

Protocol Statistician:

Behavioral and Health Outcomes Statistician:

Protocol Pathologist: Reda

### Protocol B-55/6-13 IND #122443 (olaparib), sponsored by NRG Oncology, Inc.

STUDY DRUG DRUG SUPPLY NSC#

Olaparib 747856 AstraZeneca, through the NCI

# NRG ONCOLOGY NSABP PROTOCOL B-55/BIG 6-13

**Document History** 

| | Version/Update Date | Broadcast Date |
|----------------|---------------------|-------------------|
| Amendment 7 | May 6, 2021 | 1 |
| Amendment 6 | July 27, 2018 | 1 |
| Amendment 5 | September 28, 2017 | 1 |
| Amendment 4 | July 25, 2017 | 1 |
| Amendment 3 | April 5, 2017 | April 24, 2017 |
| Amendment 2 | October 19, 2015 | February 12, 2016 |
| Amendment 1 | July 22, 2014 | September 8, 2014 |
| Activation | May 12, 2014 | July 3, 2014 |
| Pre-Activation | May 12, 2014 | June 3, 2014 |











### **Clinical Study Protocol**

Drug Substance Olaparib (AZD2281)

Study Code D081CC00006

Study Number BIG 6-13, NSABP B-55/6-13

Version 5

Date 18May2018

A randomised, double-blind, parallel group, placebo-controlled multi-centre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy

Sponsor: AstraZeneca Ab, 151 85 Södertälje, Sweden






## LIST OF OLYMPIA PROTOCOL AUTHORS

| Redacted | Medical Oncologist, Institute of Cancer Research and King's<br>College, London, UK |
|---|---|
| Redacted | Medical Oncologist, Alliance, Dana Farber Cancer Institute,<br>USA |
| Redacted | Medical Oncologist, Sheba Breast Collaborative Group (SBCG), Israel |
| Redacted | Medical Oncologist, NRG Oncology, Virginia<br>Commonwealth University Massey Cancer Center, USA |
| Redacted | Research Operations Director, Breast International Group (BIG), Belgium |
| Redacted | Medical Oncologist, Memorial Sloan-Kettering Cancer<br>Center, USA |
| Redacted | Study Statistician, NRG Oncology, USA |
| Redacted | Biostatistics Team Lead, Frontier Science (Scotland) Ltd |
| Redacted | Medical Research Fellow, Jules Bordet Institute, Belgium |
| Redacted | Head of Medical Support Team, Jules Bordet Institute,<br>Belgium |
| Redacted | Medical Oncologist, IBCSG, Hospital of Prato, Italy |
| Redacted | Medical Oncologist, Perelman School of Medicine, USA |
| Redacted | Principal Investigator/Senior Biostatistician, Frontier<br>Science and Technology Research Foundation (FSTRF),<br>Boston, MA, USA |
| Redacted | Medical Oncologist, National Cancer Institute Canada,<br>Clinical Trials Group (NCIC CTG), BC Cancer Agency,<br>Canada |
| Mediader Redacted | Senior Medical Director, Oncology Global Medicines<br>Development, AstraZeneca Gaithersburg, USA |









| Redacted | Chief Executive Officer, Breast International Group (BIG), Belgium |
|---|---|
| Redacted | Surgeon, Austrian Breast and Colorectal Cancer Group (ABCSG), Comprehensive Cancer Center Vienna, Austria |
| Redacted | Global Product Statistician, AstraZeneca Alderley Park,<br>United Kingdom |
| Redacted | Managing Director, Frontier Science (Scotland) Ltd |
| Redacted | Medical Oncologist, Chair, Breast International Group (BIG),<br>Scientific Director, Jules Bordet Institute, Belgium |
| Redacted | Medical Oncologist, Magee-Womens Hospital of UPMC,<br>NRG Oncology, USA |
| Redacted | Medical Oncologist, Breast International Group (BIG), Belgium |
| Redacted | Medical Oncologist, Center for Familial Breast and Ovarian<br>Cancer and Center of Integrated Oncology, Germany |
| Redacted | Breast Cancer Disease Area Clinical Expert, AstraZeneca<br>Alderley Park, United Kingdom |
| Redacted | Study Pathologist, Istituto Europeo di Oncologia (IEO),<br>University of Milan, Italy |
| Redacted | Gynaecologist, German BrEAST Group (GBG), Germany |
| Redacted | Senior Oncology Research Physician, AstraZeneca Alderley<br>Park, United Kingdom |
| Redacted | Senior Protocol Statistician, Frontier Science (Scotland) Ltd |
| Redacted | Senior Protocol Statistician, Frontier Science (Scotland) Ltd |
| Redacted | Global Product Statistician, AstraZeneca Gaithersburg, USA |
| Redacted | Medical Director, Breast International Group (BIG), Belgium |
| Redacted | Global Study Leader, AstraZeneca, Poland |
| Redacted | Project Manager, Breast International Group (BIG), Belgium |

#### **PROTOCOL SYNOPSIS**

A randomised, double-blind, parallel group, placebo-controlled multi-centre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy



#### Study centre(s) and number of patients planned

The study will be conducted in approximately 25 countries worldwide. Approximately 700 centres (in the US and Rest of the World countries) will be initiated to randomise approximately 1800 patients. Additional countries and sites may be added dependent on recruitment rates.

Approximately 150 randomised patients\* will be analysed for pharmacokinetic (PK) at those sites that have confirmed that they are able to collect the PK assessment samples. PK sampling will be performed in a subset of patients who sign optional PK Informed consent. PK sampling will not be done in the US.

| Study period | | Phase of development |
|------------------------------------------|---------|----------------------|
| Estimated date of first patient enrolled | Q1 2014 | III |
| Estimated date of last patient completed | 2028 | |

<sup>\*</sup> No placebo samples will be analyzed unless requested.

NCI Version Date: 05-06-2021 6(177) NSABP B-55/BIG 6-13

#### **Objectives**

#### **Primary Objective**

The primary objective is to assess the effect of adjuvant treatment with olaparib on Invasive Disease Free Survival (IDFS)

#### **Safety Objective**

To assess the safety and tolerability of adjuvant treatment with olaparib

#### **Secondary Objectives**

- 1. To assess the effect of adjuvant treatment with olaparib on overall survival (OS)
- 2. To assess the effect of adjuvant treatment with olaparib on Distant Disease Free Survival (DDFS)
- 3. To assess the effect of adjuvant treatment with olaparib on the incidence of new primary contralateral invasive breast cancer, primary contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer
- 4. To assess the effect of olaparib on patient reported outcomes using the FACIT-Fatigue and EORTC QLQ-C30 questionnaires
- 5. To assess the efficacy of olaparib in patients identified as having a deleterious or suspected deleterious variant in either of the *BRCA* genes using variants identified with current and future germline *BRCA* mutation assays (gene sequencing and large rearrangement analysis)
- 6. To determine the exposure to olaparib (in plasma) in patients receiving olaparib as adjuvant therapy.



| | Redacted |
|------|-----------|
| | Redacted |
| Reda | Redacted |
| | 1.0040.04 |

#### Study delivery model

This is a collaborative study being coordinated worldwide by the Breast International Group (BIG) in partnership with Frontier Science (FS), NRG Oncology (NCI supported National Clinical Trials Network Group) and AstraZeneca (AZ). Two versions of this protocol have been written to cover this global adjuvant breast cancer study. One protocol version covers all patients recruited outside of the US (where AZ is the sponsor) and one protocol version covers patients recruited within the US (where NRG Oncology is the sponsor). The two versions of the protocol are identical in terms of study objectives and scientific content and only differ in logistical content appropriate for the country(ies) they cover (i.e. drug distribution, mechanisms for SAE reporting during the study, etc.). Based on current recruitment rates, it is expected that approximately 230 patients will be randomised under the US protocol and approximately 1570 patients will be randomised under the Rest of the World protocol.

The trial will use one randomisation system and report as one single study. The initial collection of the patients' data will be done using two databases (one for the US patients and one for all other patients outside of the US). The two databases will be set up using the same standards and eCRFs to ensure consistency in the data collection. The data from both databases will be combined into a single consolidated database at regular, pre-specified intervals. All study endpoints as well as reports for periodic review by the Independent Data Monitoring Committee

(IDMC) will be analysed and reported from the single combined reporting database held by Frontier Science on behalf of BIG.

#### Study design

This is a randomised, double-blind, parallel group, placebo-controlled multi-centre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy.

Patients will be randomised in a 1:1 ratio to either olaparib or placebo. Randomisation will be stratified by hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC), by prior neoadjuvant versus adjuvant chemotherapy, and prior platinum use for breast cancer (yes versus no).

Eligible patients with deleterious or suspected deleterious *gBRCA* mutations and high risk HER2 negative breast cancer should be randomised in the trial ideally within a maximum of 8 weeks of completing their last treatment modality (chemotherapy and definitive local or locoregional treatment), but in no case longer than 12 weeks. Randomised patients will receive study treatment for up to a maximum of 12 months. All patients will have safety assessments every 2 weeks during the first month, every 4 weeks for the following 5 months (up to week 24) and 3 monthly for the remaining 6 months of study treatment plus 30 days after its discontinuation. All randomised patients will have clinical assessment visits for approximately 10 years following their randomisation into the study, or until an IDFS endpoint due to a breast cancer related distant relapse, whichever comes first. They then enter the annual survival follow-up phase of the trial, which will continue until 10 years after the last patient is randomised. No clinic visits will be required during the survival follow-up phase; information may be collected via telephone, medical records or death registries.

#### **Target patient population**

Patients eligible for the trial are those with a deleterious or suspected deleterious germline *BRCA* mutation (defined by local or central Myriad testing) with high risk HER2 negative primary breast cancer who have completed definitive local treatment, and neoadjuvant or adjuvant chemotherapy. Definitions of high risk HER2 negative patients are provided below.

- 1. For patients who underwent initial surgery and received adjuvant chemotherapy
  - TNBC patients must have been axillary node-positive-(≥pN1, any tumour size) or axillary node negative (pN0) with invasive primary tumour pathological size
     2 cm (≥pT2).
  - ER and/or PgR positive/HER2 negative patients must have had ≥ 4 pathologically confirmed positive lymph nodes.

- 2. For patients who underwent neoadjuvant chemotherapy followed by surgery
  - TNBC patients must have residual invasive breast cancer in the breast and/or resected lymph nodes (non pCR)
  - ER and/or PgR positive/HER2 negative patients must have residual invasive cancer in the breast and/or the resected lymph nodes (non pCR) AND a CPS&EG score ≥3. (Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS) a disease scoring system). Instructions how to calculate CPS&EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix H.

#### Germline BRCA1 and BRCA2 (gBRCA) testing

Local *gBRCA* testing results, if available, can be used for establishing eligibility. If local *gBRCA* testing results are not available, central testing will be provided for those patients who otherwise appear to be eligible. Irrespective of the availability of local *gBRCA* testing results, all patients must provide a sample for central *gBRCA* testing.

## Central tumour analyses (e.g. somatic *BRCA1/2* functional status, ER/PgR and HER2 status)

Archival tumour samples must be provided for all patients.

For adjuvant patients, this refers to the surgical specimen; for neoadjuvant patients, both the pretreatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required.

#### Study treatment, dosage and mode of administration

AstraZeneca's Pharmaceutical Development, R&D Supply Chain will supply olaparib and matching placebo as green film-coated tablets to the Pharmaceutical Management Branch, Division of Cancer Therapy and Diagnosis, National Cancer Institute.

Patients will be randomised in a 1:1 ratio to one of the following treatments:

- 12 months treatment with olaparib tablets p.o. 300 mg twice daily (two 150 mg tablets in the morning and two 150 mg tablets in the evening)
- 12 months treatment with matching placebo tablets p.o. twice daily (two tablets in the morning and two tablets in the evening)

#### **Stratification**

Patients will be stratified at randomisation by the following baseline factors:

- Hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC)
   NOTE: In cases of multifocal, multicentric or synchronous bilateral invasive disease, stratification is based on the status of the lesion considered at highest risk (at the investigator's discretion) that was used to determine eligibility.
- Neoadjuvant versus adjuvant chemotherapy
- Platinum therapy for current breast cancer: Yes/No

Within this study, patients will not be provided with olaparib post discontinuation of study treatment. Patients and investigators will not be routinely unblinded to study treatment prior to the final overall survival (OS) analysis. Unblinding is allowed only in the case of compelling medical or safety reasons (Section 5.4.2).

#### **Outcome(s):**

- Primary outcome
  - Invasive Disease Free Survival (IDFS)
- Secondary outcomes
  - Overall Survival (OS)
  - Distant Disease Free Survival (DDFS)
  - New primary contralateral breast cancers (invasive and non-invasive), new primary ovarian cancer, new primary fallopian tube cancer, and new primary peritoneal cancers in patients at risk for these events
  - FACIT-Fatigue symptom scale score and EORTC-QLQ-C30 global health status, functional, and symptoms scales/items scores
  - IDFS, DDFS and OS based on patients with gBRCA mutations confirmed by the central test (only required if population differs from the ITT (intention to treat) population)
  - Pharmacokinetic analysis
- Safety outcomes
  - Adverse Events (AE), physical examination, vital signs including blood pressure
     (BP), pulse, and laboratory findings including clinical chemistry and haematology



#### **Statistical methods**

The primary endpoint of the study is IDFS and patients will be randomised 1:1 to either olaparib 300 mg b.i.d. (twice daily) or matching placebo.

Approximately 1800 patients will be randomised into the study. If the true hazard ratio for the comparison of olaparib versus placebo in terms of IDFS is 0.7 then with 330 events, the analysis of IDFS will have 90% power to demonstrate a statistically significant difference in IDFS, assuming a 2-sided 5% significance level. It is estimated the study will take approximately 5 years to complete recruitment of approximately 1800 patients. The primary analysis will be triggered by the occurrence of 330 IDFS events (required for overall 90% power to detect a HR of 0.7). Assuming a nonuniform recruitment, the primary analysis is estimated to occur approximately 6 years from the start of randomisation.

An interim analysis for superiority will be performed once a minimum of 165 IDFS events have been observed from the first 900 patients recruited. It is estimated that this analysis will occur approximately 5.3 years after the first patient is randomised. Consideration of futility will also be made at the time of interim analysis.

Safety data will be summarised descriptively in terms of AEs, vital signs, clinical chemistry & haematology and physical exam and will include all patients who received at least one dose of olaparib or placebo.

Patient reported outcomes and health related quality of life (HRQoL) will be assessed through the planned correlative study using the FACIT-Fatigue and the EORTC QLQ-C30 questionnaires.

An analysis of IDFS, DDFS and OS will be conducted based on patients with *gBRCA* mutations confirmed by the central test, if this population differs from the primary ITT population. Similar sensitivity analyses will be performed based on ER and/or PgR positive/HER2 negative and TNBC subsets as defined by the central laboratory testing.

Full details of all the statistical analyses will be documented in the SAP. Version 1.0 of the SAP will be prepared prior to first subject in (FSI).

#### Pharmacokinetic analysis

The plasma concentration-time data will be analysed by non-linear mixed effects modelling in order to evaluate the pharmacokinetic characteristics of olaparib, quantify variability in the pharmacokinetics, identify demographic or pathophysiological covariates, which may explain the observed variability and explore exposure-response relationships.

| TABLE | OF CONTENTS | PAGE |
|---|---|---|
| | NSABP PROTOCOL B-55/BIG 6-13 | 1 |
| | LIST OF OLYMPIA PROTOCOL AUTHORS | 4 |
| | PROTOCOL SYNOPSIS | 6 |
| | INFORMATION RESOURCES | 20 |
| | CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION | 22 |
| | LIST OF ABBREVIATIONS AND DEFINITION OF TERMS | 23 |
| 1. | INTRODUCTION | 28 |
| 1.1 | Background | 28 |
| 1.1.1 | Breast cancer and its treatment | 28 |
| 1.1.2 | Triple Negative Breast Cancer (TNBC) | 29 |
| 1.1.3 | Adjuvant chemotherapy for TNBC | 29 |
| 1.1.4 | Neoadjuvant chemotherapy for TNBC | 29 |
| 1.1.5 | ER/PgR positive HER2 negative breast cancer with germline BRCA | 20 |
| 1.1.6 | mutations | 30 |
| 11110 | cancer | 31 |
| 1.1.7 | Pre-clinical experience | |
| 1.1.8 | Toxicology and safety pharmacology summary | |
| 1.1.9 | Clinical experience | |
| 1.1.9.1 | Olaparib monotherapy studies in breast cancer patients | |
| 1.2 | Research hypothesis | 33 |
| 1.3 | Rationale for conducting this study | 34 |
| 1.3.1 | Rationale for central BRCA mutation test at Myriad Genetics, Inc | |
| 1.4 | Benefit/risk and ethical assessment | 35 |
| 2. | STUDY OBJECTIVES | 40 |
| 2.1 | Primary objective | 40 |
| 2.2 | Secondary objectives | 40 |
| 2.3 | Safety objective | 41 |
| Redacted | | 41 |
| 3. | STUDY PLAN AND PROCEDURES | 42 |
| 3.1 | Overall study design, flow chart and study schedules | 42 |
| 3.2 | Rationale for study design, doses and control groups | 55 |
| 3.2.1 | Rationale for study design. | |
| 3.2.2 | Rationale for patient reported outcomes | |
| 3.2.3 | Study Population | |

| 4. | PATIENT SELECTION CRITERIA | 58 |
|---|---|---|
| 4.1 | Inclusion criteria | 58 |
| 4.2 | Exclusion criteria | 62 |
| 5. | STUDY CONDUCT | 64 |
| 5.1<br>5.1.1<br>5.1.2 | Restrictions during the study Meals and dietary restrictions Contraception | 64 |
| 5.2<br>5.2.1<br>5.2.2<br>5.2.2.1<br>5.2.2.2<br>5.2.2.3<br>5.2.2.4<br>5.2.2.5<br>5.2.3<br>5.2.4 | Patient enrolment and randomisation and initiation of study treatment. CTEP registration procedures CTSU registration procedures IRB approval Downloading site registration documents Requirements for B-55/6-13 site registration Submitting regulatory documents Checking your site's registration status Procedures for randomisation Oncology Patient Enrollment Network (OPEN) | 65 66 67 67 67 68 |
| 5.3 | Procedures for handling patients incorrectly enrolled or randomised or initiated on study treatment | |
| 5.4<br>5.4.1<br>5.4.2<br>5.4.3 | Blinding and procedures for unblinding the study Methods for ensuring blinding Methods for unblinding individual patients Procedures for unblinding | 70<br>70 |
| 5.5<br>5.5.1<br>5.5.2<br>5.5.2.1<br>5.5.3 | Treatments Identity of study treatment Doses and treatment regimens Olaparib and matching placebo (study treatment) Olaparib/Placebo | 71<br>71<br>71 |
| 5.5.3.1<br>5.5.4<br>5.5.5<br>5.5.6 | Obtaining an Investigator's Brochure Procurement of olaparib (IND #122443, NSC #747856)/placebo Special ordering procedures for patients requiring a dose reduction | 75<br>75<br>76 |
| 5.5.7<br>5.5.8<br>5.5.9<br>5.5.10 | Agent inventory records Useful Links and Contacts Transfer of olaparib/placebo Return of olaparib/placebo | 76<br>76 |
| 5.5.11<br>5.5.12<br>5.5.12.1<br>5.5.12.2 | Labelling | 77<br>78<br>78 |
| 5.5.12.3<br>5.5.12.4<br>5.5.12.5 | Renal impairment | 82<br>82 |

| 5.5.12.6<br>5.5.12.7 | Management of nausea and vomiting Interruptions for intercurrent non-toxicity related events | |
|---|---|---|
| | - | |
| 5.6<br>5.6.1 | Concomitant and subsequent treatment(s) | 8 <i>3</i> |
| 5.6.2 | Restricted concomitant medications | |
| 5.6.3 | Anti-emetics/Anti-diarrheals | |
| 5.6.4 | Live virus and bacterial vaccines | |
| 5.7<br>5.7.1 | Treatment compliance | |
| 5.8<br>5.8.1 | Discontinuation of study treatment Procedures for discontinuation of a patient from study treatment | |
| 5.9 | Withdrawal from study | |
| 6. | COLLECTION OF STUDY VARIABLES | |
| 6.1 | Recording of data | |
| 6.1.1 | Instructions for completion of B-55/6-13 forms and materials | 90 |
| 6.1.2 | Instructions for submission of B-55/6-13 data, forms, and materials | |
| 6.1.3 | Data monitoring for CTEP | |
| 6.2 | Study procedures | 91 |
| 6.2.1 | Screening procedures | |
| 6.2.2 | On-treatment assessments | 94 |
| 6.2.3 | Efficacy follow-up assessments | 95 |
| 6.2.4 | Safety follow-up assessments 30 days after last dose of olaparib/placebo | |
| 6.2.5 | Patient management post-primary analysis | |
| 6.2.6 | Patient management post-final analysis | |
| 6.3 | Efficacy | |
| 6.3.1 | Tumour evaluation | 97 |
| 6.4 | Safety | 98 |
| 6.4.1 | Investigational agents | 98 |
| 6.4.2 | Commercial agents | |
| 6.4.3 | Double-blind study drug | |
| 6.4.4 | Adverse event characteristics | |
| 6.4.5 | Definition of adverse events (AE) | |
| 6.4.6<br>6.4.7 | Definitions of serious adverse event (SAE) | |
| 6.4.8 | Expedited reporting of adverse events | |
| 6.4.8.1 | Expedited reporting of adverse events Expedited reporting methods | |
| 6.4.8.2 | Protocol-specific expedited reporting requirements | |
| 6.4.9 | Recording of adverse events | |
| 6.4.10 | Reporting of serious adverse events | |
| 6.4.11 | Laboratory safety assessment | |
| 6.4.11.1 | Full haematology assessments for safety | 109 |
| 6.4.11.2 | Coagulation | |
| 6.4.11.3 | Clinical chemistry assessments for safety | 109 |

| 6.4.11.4 | Urinalysis | 11( | ) |
|---|---|---|---|
| 6.4.11.5 | Bone marrow or blood cytogenetic samples | 110 | ) |
| 6.4.12 | Physical examination. | | |
| 6.4.13 | ECG | | |
| 6.4.13.1 | Resting 12-lead ECG | | |
| 6.4.14 | Vital signs | | |
| 6.4.14.1 | Pulse and blood pressure | | |
| 6.4.14.2<br>6.4.15 | Body temperature | | |
| 6.4.15.1 | Other safety assessments | | |
| | Serum or urine pregnancy test | | |
| 6.5 | Patient reported outcomes (PRO) | | |
| 6.5.1 | FACIT-Fatigue | | |
| 6.5.2 | EORTC QLQ-C30 | | |
| 6.5.3 | Administration of PRO questionnaires | | |
| 6.5.4 | Reimbursement | | |
| 6.6 | Biomarkers | | |
| 6.6.1 | Biomarker samples | | |
| 6.6.2 | Collection of blood sample for Myriad germline <i>BRCA1</i> and <i>BRCA2</i> testing | 113 | , |
| 6.6.2.1 | Collection of a blood sample for assessment of current and future BRCA | 111 | _ |
| ((2 | mutation assay(s) | | |
| 6.6.3<br>6.6.4 | Redacted | 116 | ) |
| 0.0.4 | Redacted Redacted | 114 | |
| | | 11( | , |
| 665 | Redacted | | |
| 6.6.5 | Redacted Redacted | 117 | 7 |
| | Redacted | 117<br>117 | |
| 6.6.6 | Redacted | 117 | 7 |
| 6.6.6<br>6.7 | Redacted | <ul><li>117</li><li>117</li></ul> | 7 |
| 6.6.6<br>6.7<br>6.7.1 | Redacted | 117<br>117<br>117 | 7<br>7 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8 | Redacted | <ul><li>117</li><li>117</li><li>117</li><li>118</li></ul> | 7 7 3 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1 | Redacted Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) | 117<br>117<br>117<br>118<br>118 | 7 7 3 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2 | Redacted Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) Collection of samples | 117<br>117<br>118<br>118<br>118 | 7 7 3 3 3 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3 | Redacted Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) Collection of samples Determination of drug concentration | 117<br>117<br>118<br>118<br>118 | 7 7 3 3 3 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3<br>6.9 | Redacted Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) Collection of samples Determination of drug concentration Health economics | 113<br>113<br>113<br>118<br>118<br>119 | 7 7 3 3 3 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3<br>6.9 | Redacted Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) Collection of samples Determination of drug concentration | 113<br>113<br>113<br>118<br>118<br>119 | 7 7 3 3 3 |
| 6.7.1 | Redacted Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) Collection of samples Determination of drug concentration Health economics | 117<br>117<br>118<br>118<br>118<br>119<br>119 | 7 7 3 3 9 9 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3<br>6.9<br>6.9.1 | Redacted Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) Collection of samples Determination of drug concentration Health economics Resource use (serious adverse events) | 113<br>113<br>118<br>118<br>118<br>119<br>119 | 7 7 8 8 9 9 9 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3<br>6.9<br>6.9.1 | Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) Collection of samples Determination of drug concentration Health economics Resource use (serious adverse events) BIOLOGICAL SAMPLING PROCEDURES Volume of blood. | 113<br>113<br>118<br>118<br>118<br>119<br>119<br>119 | 7 7 7 8 8 8 9 9 9 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3<br>6.9<br>6.9.1<br>7. | Redacted Redacted Pharmacokinetics (Optional) | 113<br>113<br>118<br>118<br>118<br>119<br>119<br>119<br>120<br>120 | 7 7 7 8 8 8 9 9 9 9 9 9 9 9 9 9 9 9 9 9 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3<br>6.9<br>6.9.1<br>7. | Redacted Redacted Pharmacokinetics (Optional) | 113<br>113<br>118<br>118<br>118<br>119<br>119<br>119<br>120<br>120 | 7 7 7 8 8 8 9 9 9 9 9 9 9 9 9 9 9 9 9 9 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3<br>6.9<br>6.9.1<br>7.<br>7.1<br>7.2<br>7.2.1 | Redacted Redacted Pharmacokinetics (Optional) | 113<br>113<br>118<br>118<br>119<br>119<br>119<br>120<br>120<br>121 | 7 7 3 3 3 9 9 1 |
| 6.6.6<br>6.7<br>6.7.1<br>6.8<br>6.8.1<br>6.8.2<br>6.8.3<br>6.9<br>6.9.1<br>7.<br>7.1<br>7.2<br>7.2.1<br>7.2.2 | Redacted Redacted Redacted Pharmacokinetics (Optional) Pharmacokinetic samples (Subset of patients) Collection of samples Determination of drug concentration Health economics Resource use (serious adverse events) BIOLOGICAL SAMPLING PROCEDURES Volume of blood Handling, storage and destruction of biological samples. Pharmacogenetic samples Pharmacokinetic samples | 113<br>113<br>118<br>118<br>118<br>119<br>119<br>120<br>120<br>121 | 7 7 7 8 8 8 9 9 9 1 1 1 |

| 8. | ETHICAL AND REGULATORY REQUIREMENTS | 123 |
|---|---|---|
| 8.1 | Ethical conduct of the study | 123 |
| 8.2 | Patient data protection | 123 |
| 8.3 | Ethics and regulatory review | 124 |
| 8.4 | Informed consent | 124 |
| 8.5 | Changes to the protocol and informed consent form | 125 |
| 8.6 | Audits and inspections. | 125 |
| 9. | STUDY MANAGEMENT | 126 |
| 9.1 | Pre-study activities | 126 |
| 9.2 | Training of study site personnel | 126 |
| 9.3 | Monitoring of the study | 126 |
| 9.4 | Study timetable and end of study | 127 |
| 10. | DATA MANAGEMENT | 127 |
| 11. | EVALUATION AND CALCULATION OF VARIABLES | 128 |
| 11.1<br>11.1.1<br>11.1.2<br>11.1.2.1<br>11.1.2.2<br>11.1.2.3 | Calculation or derivation of efficacy variable(s) | 128<br>129<br>129<br>129 |
| 11.2<br>11.2.1 | Calculation or derivation of safety variable(s) | 131 |
| 11.3 | Calculation or derivation of patient reported outcome variables | 131 |
| 11.4 | Calculation or derivation of pharmacokinetic variables | 131 |
| 11.5 | Calculation or derivation of pharmacodynamic variable(s) - not applicable | 131 |
| 11.6 | Calculation or derivation of Redacted variables | 131 |
| 11.7 | Calculation or derivation of health economic variables –not applicable | 131 |
| 12. | STATISTICAL METHODS AND SAMPLE SIZE DETERMINATION | 131 |
| 12.1<br>12.1.1<br>12.1.2<br>12.1.3 | Description of analysis sets Full analysis set Safety analysis set PK Analysis set | 132<br>132 |
| 12.2<br>12.2.1 | Methods of statistical analysis | |

| 12.2.1.1 | Primary analysis | |
|---|---|---|
| 12.2.1.2<br>12.2.1.3 | Sensitivity analysis | |
| 12.2.1.3 | Subgroup analysis Analysis of interaction | |
| 12.2.1.4 | Analysis of secondary endpoints | |
| 12.2.3 | Analysis of patient reported outcomes | |
| 12.2.3.1 | Hypotheses and objectives | |
| 12.2.3.2 | Statistical considerations for patient reported outcomes | 139 |
| 12.2.3.3 | Pharmacokinetic analysis | |
| 12.2.4 | Multiplicity strategy for primary and key secondary endpoints | 141 |
| 12.2.5<br>12.2.6 | | |
| 12.2.7 | Interim analysis | |
| 12.2.7 | Issues relating to racial and ethnic differences in the U.S | |
| 12.3 | Independent data monitoring committee | |
| 13. | IMPORTANT MEDICAL PROCEDURES TO BE FOLLOWED BY THE INVESTIGATOR | 149 |
| 13.1 | Medical emergencies and contacts | 149 |
| 13.2 | Overdose | 150 |
| 13.3 | Pregnancy | 150 |
| 13.3.1<br>13.3.2 | Maternal exposure Expedited reporting of pregnancy, pregnancy loss, and death neonatal | 150 |
| 13.3.2 | occurring during study therapy | 151 |
| 13.3.3 | Paternal exposure | |
| 14. | LIST OF REFERENCES | 152 |
| LIST O | F TABLES | |
| Table 1 | Study Schedule - Screening (PART 1 and PART 2) | 46 |
| Table 2 | Study Schedule – On treatment (Year 1) | 49 |
| Table 3 | Study Schedule - Follow-up Visits (Year 2 onwards) | 53 |
| Table 4 | Identity of study treatment | 71 |
| Table 5 | Study treatment doses and treatment regimens | |
| Table 6 | Olaparib/placebo dose levels | 79 |
| Table 7 | Mandatory treatment for hematologic toxicity and treatment guidance for other olaparib/placebo toxicities | 80 |
| Table 8 | Dose reduction for study treatment to manage moderate renal impairment | 81 |
| Table 9 | Dose reduction for study treatment with concurrent use of a strong or | 25 |
| | moderate CYP3A inhibitor | 82 |

| Table 10 | Restricted concomitant medications. | 85 |
|---|---|---|
| Table 11 | Late Phase 2 and Phase 3 Studies: Expedited reporting requirements for adverse events that occur on studies under an IND within 30 days of the last administration of the investigational agent (olaparib/placebo) <sup>1</sup> | 102 |
| Table 12 | Samples for Biomarker Research | |
| | Volume of blood to be drawn from each patient | |
| | Summary of Outcome Variables and Analysis Populations | |
| | Summary of 2-sided significance levels and total alpha spend across the endpoints and analyses | |
| Table 16 | Actual accrual between June 2014 and February 2018 | 146 |
| Table 17 | Expected racial and ethnic composition of NSABP B-55/BIG 6-13 | 147 |
| Table 18 | Point assignments for the CPS + EG staging system | 176 |
| LIST O | FFIGURES | |
| Figure 1 | Study Flow Chart | 44 |
| Figure 2 | Screening Plan | 45 |
| Figure 3 | Multiple testing procedure | 142 |
| LIST O | FAPPENDICES | |
| Appendix | A Additional Safety Information | 160 |
| | B International Airline Transportation Association (IATA) 6.2 Guidance | |
| 11 | Document | 162 |
| Redacted | Redacted | 163 |
| Appendix | D Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law | |
| Appendix | E Acceptable Birth Control Methods | 171 |
| Appendix | F ECOG Performance Status | 172 |
| Appendix | G Patient Reported Outcomes (FACIT-Fatigue, EORTC QLQ-C30) | 173 |
| Appendix | H CPS & EG Score | 176 |

## INFORMATION RESOURCES

| NRG Oncology | | |
|---|---|---|
| Redacted | | |
| NRG Oncology | Redacted | Phone: Redacted |
| NRG Oncology<br>Statistics and Data<br>Management Center<br>(SDMC) | Redacted | Phone: Redacted Fax: Redacted (General office fax) |
| Questions/problems<br>regarding IRB review &<br>informed consent | NRG Oncology Redacted Department of Regulatory Affairs | Phone: Redacted E-mail: Redacted |
| Submission of IRB approval | Redacted | Submit to the CTSU via the Regulatory Submission Portal Redacted |
| Questions concerning eligibility and clinical aspects of the trial | NRG Oncology Redacted Clinical Coordinating Department | Phone: Redacted E-mail: Redacted |
| Study entry information (see <u>Section</u> 5.2) | NRG Oncology SDMC<br>Patient Entry Coordinator | Phone: Redacted |
| Request for kits for<br>tumor and blood sample<br>collections | Refer to the B-55/6-13 Pathology and<br>B-55 Web page of the CTSU Member | Correlative Science Instructions in the Web site at Redacted |
| Arrangement for return of blocks that are not to be stored | NRG Oncology<br>Biospecimen Bank Redacted | Phone: Redacted E-mail: Redacted |
| | NRG Oncology SDMC | Phone: Redacted Fax: Redacted |
| Questions concerning drug orders, shipments, transfers, and returns of olaparib (see Section 5.5) | For mail (USPS): Pharmaceutical Management Branch, CTEP, DCTD Redacted For express courier: Pharmaceutical Management Branch, CTEP, DCTD Redacted | Phone: Redacted Fax: Redacted E-mail: Redacted |

Continued on next page.

## INFORMATION RESOURCES (continued)

| Requests for unblinding<br>(including 24-hour<br>emergency unblinding) | NRG Oncology SDMC | Phone: Redacted |
|---|---|---|
| Questions concerning expedited adverse event reporting (see Section 6.4.8) | NRG Oncology SDMC<br>B-55/6-13 AE Reporting Nurse | Phone: Redacted Fax: Redacted E-mail: Redacted |
| Submission of patient-<br>completed<br>questionnaires (see<br><u>Section</u> <u>6.1.2</u> ) | NRG Oncology SDMC<br>B-55/6-13 Data Manager | Phone: Redacted Fax: Redacted Redacted Redacted |
| Submission of data<br>forms/questions<br>concerning data<br>management and<br>Medidata Rave | NRG Oncology SDMC<br>B-55/6-13 Data Manager | Phone Redacted Redacted |

# CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| For regulatory requirements: | For patient enrollments: | For study data submission: |
|---|---|---|
| Regulatory documentation must be submitted to the CTSU via the Regulatory Submission Portal: | Please refer to the patient | Data collection for this study |
| Regulatory Submission Portal (Sign in at Redacted and select the Regulatory Submission sub-tab under the | enrollment section of the protocol for instructions on using Oncology Patient Enrollment Network (OPEN), | will be done exclusively through Medidata Rave. Refer to Section 6.1.2 for further instructions. |
| Regulatory tab.) Institutions with patients waiting that are unable to use the Portal should alert the | which can be accessed at Redacted OPEN SYSTEM/ or Redacted | Submit patient-completed questionnaires to the NRG Oncology as directed on the worksheet. |
| CTSU Regulatory Office immediately at Redacted to receive further instruction and support. | Contact the CTSU Help Desk with any OPEN-related questions at Redacted | Do <u>not</u> submit study data or forms to CTSU Data Operations. Do <u>not</u> copy the CTSU on data submission. |
| Contact the CTSU Regulatory Help Desk at Redacted for regulatory assistance. | | |
| downloaded from the protocol-<br>Redacted Access to<br>Therapy and Evaluation Progra | study protocol and all suppor<br>specific Web page of the CTSU<br>o the CTSU Members' website is<br>m-Identity and Access Managen<br>with CTEP-IAM username and | Member Web site located at s managed through the Cancer nent (CTEP-IAM) registration |
| For clinical questions (i.e., pa<br>Coordinating Department at NE<br>Redacted | tient eligibility and treatment-<br>RG Oncology at Redacted 7 | related), contact the Clinical or by e-mail at |
| For non-clinical questions (i.e submission) contact the CTSU | e., unrelated to patient eligibilit<br>Help Desk by phone or email: | y, treatment, or clinical data |
| CTSU General Information Lin<br>correspondence will be triaged | ne – Redacted or Redacted to the appropriate CTSU represe | |
| The CTSU Web site is located | atRedacted | |

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

The following abbreviations and special terms are used in this study Clinical Study Protocol.

| Abbreviation or special term | Explanation |
|---|---|
| AE | Adverse event (see definition in <u>Section</u> <u>6.4.5</u> ) |
| AESI | Adverse event of special interest |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AML | Acute Myeloid Leukaemia |
| ANC | Absolute neutrophil count |
| APTT | Activated Partial Thromboblastin Time |
| ASCO | American society of Clinical Oncology |
| AST | Aspartate aminotransferase |
| AUC | Area Under Curve |
| b.i.d | Twice daily |
| BP | Blood Pressure |
| BRCA | Breast cancer susceptibility gene |
| BUN | Blood Urea Nitrogen |
| CA-125 | Cancer antigen-125 |
| cfDNA | Circulating free DNA |
| СНО | Chinese hamster ovary |
| CI | Confidence Interval |
| Cmax <sub>ss</sub> | Maximum concentration at steady state |
| Cmin <sub>ss</sub> | Minimum concentration at steady state |
| CNS | Central Nervous System |
| CPS&EG | Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS) - a disease scoring system |
| CR | Complete Response |
| CRF (eCRF) | Case Report Form (electronic/paper) |
| CRO | Contract Research Organisation |
| CSA | Clinical Study Agreement |
| CSR | Clinical Study Report |
| CT | Computerised Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |

| Abbreviation or special term | Explanation |
|---|---|
| CTEP | Cancer Therapy Evaluation Program |
| CTEP-AERS | CTEP Adverse Event Reporting System |
| CTEP-IAM | CTEP Identity and Access Management |
| CTSU | Cancer Trials Support Unit |
| DAE | Discontinuation of study treatment due to Adverse Event |
| DCIS | Ductal carcinoma in situ |
| DCO | Data cut off |
| DCTD | Division of Cancer Treatment and Diagnosis |
| DDFS | Distant disease free survival |
| DFS | Disease free survival |
| DNA | Deoxyribonucleic acid |
| DSB | Double strand break |
| DUS | Disease under Study |
| EC | Ethics Committee, synonymous to Institutional Review Board (IRB) and Independent Ethics Committee (IEC) |
| ECG | Electrocardiogram |
| ECOG performance status | Eastern Cooperative Oncology Group performance status using scales and criteria to assess how a patient's disease is progressing |
| EORTC QLQ-C30 | The European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire-Core questions 30 |
| ER | Estrogen receptor |
| ESMO | European Society for Medical Oncology |
| ESTRO | European Society for Radiation and Oncology |
| FACIT-Fatigue | Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue<br>Measurement questionnaire |
| FAS | Full Analysis Set |
| FFPE | Formalin Fixed Paraffin Embedded |
| FSH | Follicle Stimulating Hormone |
| gBRCA mutation or gBRCAm | The term "gBRCA mutation" is used to refer to a germline BRCA1 or BRCA2 mutation classified as "deleterious" or "suspected deleterious" in accordance with the American College of Medical Genetics and Genomics recommendations for standards for interpretation and reporting of sequence variants |
| GCP | Good Clinical Practice |

| Abbreviation or special term | Explanation |
|---|---|
| GMP | Good Manufacturing Practice |
| HDPE | High Density Polyethylene |
| HER2 | Human Epidermal Growth Factor Receptor 2 |
| Hgb | Hemoglobin |
| HR | Hazard Ratio |
| HRD | Homologous Recombination Deficiency |
| HRQoL | Health Related Quality of Life |
| IAM | Identity and Access Management |
| IB | Investigators Brochure |
| ICH | International Conference on Harmonisation |
| International<br>Co-ordinating<br>investigator | If a study is conducted in several countries, the International Co-ordinating Investigator is the Investigator co-ordinating the investigators and/or activities internationally. |
| IDFS | Invasive Disease-free Survival |
| IDMC | Independent Data Monitoring Committee |
| IHC | Immunohistochemistry |
| IIBTR | Ipsilateral invasive breast tumour recurrence |
| INR | International Normalised Ratio |
| IPCW | Inverse Probability of Censoring Weighting |
| IRB | Institutional Review Board |
| ISH | In Situ Hybridisation (includes FISH, DISH, CISH) |
| ISS | Investigator Sponsored Study |
| ITT | Intention To Treat |
| IVRS | Interactive Voice Response System |
| IWRS | Interactive Web Response System |
| KM | Kaplan-Meier |
| LDH | Lactic Dehydrogenase |
| LIMS | Laboratory Information Management System |
| LLOQ | Lower Limit of Quantification |
| LSI | Last Subject in |
| LSLV | Last Subject Last Visit |
| MCH | Mean Cell Haemoglobin |
| MCHC | Mean Cell Haemoglobin Concentration |

| Abbreviation or special term | Explanation |
|---|---|
| MCV | Mean Cell Volume |
| MDS | Myelodysplastic Syndrome |
| MMRM | Mixed Model for Repeated Measures |
| MRI | Magnetic Resonance Image |
| MTD | Maximum Tolerated Dose |
| MTP | Multiple testing procedure |
| NCCN | National Comprehensive Cancer Network |
| NCI | National Cancer Institute |
| NCTN | National Clinical Trials Network |
| NSABP | National Surgical Adjuvant Breast and Bowel Project |
| NSC | National Service Center |
| NSCLC | None Small cell lung cancer |
| OAE | Other Significant Adverse Event (see definition in <u>Section 11.2.1</u> ) |
| OD | Once Daily |
| OPEN | Oncology Patient Enrollment Network |
| OR | Objective Response |
| ORR | Objective Response Rate |
| OS | Overall survival |
| PARP | Polyadenosine 5'diphosphoribase [poly (ADP ribose)] polymerisation |
| pCR | Pathological Complete Response |
| PD | Pharmacodynamics |
| PFS | Progression Free Survival |
| PFS2 | Time to second progression |
| PgR | Progesterone receptor |
| PGx | Pharmacogenetic research |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| PMB | Pharmaceutical Management Branch |
| PO | Per Os (by mouth) |
| PRO | Patient Reported Outcome |
| QOL | Quality of Life |

| Abbreviation or special term | Explanation |
|---|---|
| QT/QTc | A measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (c indicates the corrected value for this time period) |
| RBC | Red Blood Cells |
| RECIST | Response Evaluation Criteira in Solid tumours. This study will use modified RECIST version 1.1. |
| REML | Restricted Maximum Likelihood |
| RPSFT | Rank Preserving Structural Failure Time |
| RSS | Regulatory Support System |
| SAE | Serious adverse event (see definition in <u>Section</u> <u>6.4.6</u> ). |
| SAP | Statistical Analysis Plan |
| SCLC | Small Cell Lung Cancer |
| SD | Stable Disease |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic-pyruvic transaminase |
| SNB | Sentinel Node Biopsy |
| SSB | Single Strand Break |
| STEEP | Standardised Terms for Efficacy Endpoints |
| Study treatment | Study treatment is the treatment to which patient was randomised. In this study it is either olaparib or placebo |
| TN1-3 | TNM classification. Axillary node positive disease regardless of the tumour size |
| TNBC | Triple negative breast cancer |
| TPC | Chemotherapy of physician's choice |
| ULN | Upper Limit of Normal |
| WBC | White Blood Cells |
| WBDC | Web Based Data Capture |
| Wt | Wildtype (patients without evidence of <i>BRCA1</i> or <i>BRCA2</i> deleterious or suspected deleterious mutations) |

#### 1. INTRODUCTION

#### 1.1 Background

#### 1.1.1 Breast cancer and its treatment

Breast cancer is a life-threatening disease and is the second leading cause of cancer death among women. In 2013, an estimated 232,340 new cases of invasive breast cancer were expected to be diagnosed among US women, and approximately 39,620 women were expected to die from breast cancer (<u>American Cancer Society 2013</u>). In the European Community, the estimated age adjusted annual incidence in 2008 was 88.4/100 000 and the mortality 24.3/100 000 (<u>Aebi et al 2011</u>).

Approximately 5% of breast cancers are associated with a mutation in the *BRCA1* and/or *BRCA2* gene with approximately 3% associated with the *BRCA1* gene (generally presenting with TNBC phenotype) and approximately 2% associated with the *BRCA2* gene (generally ER/PgR positive phenotype). In the general population, *BRCA* mutation carriers have an increased relative risk of breast cancer. The presence of *BRCA1* mutations is associated with a lifetime risk of breast cancer of 60 to 70% and a lifetime risk of ovarian cancer of 20 to 45% (Antoniou et al 2003). *BRCA2* mutations are associated with lifetime risk of breast cancer of 40 to 60% in women and 5 to 10% in men and a lifetime risk of ovarian cancer of 10 to 20%. Rare individuals carry deleterious mutations in both *BRCA1* and *BRCA2* genes.

In breast cancer, there are differences between *BRCA1* and *BRCA2* mutation carriers. Approximately 70% of breast cancer patients with *BRCA1* mutations present as triple negative breast cancer (TNBC). In contrast, patients carrying mutations in the *BRCA2* gene are more likely to be positive for expression of the estrogen receptor in their breast cancer while approximately 20% will have triple negative cancers (Mavaddat et al 2012).

Although there are phenotypic differences in breast cancers resulting from *BRCA1* or *BRCA2* mutations, their important commonality is that mutations in either gene result in tumours that are deficient in homologous recombination, making both appropriate for treatment with polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerisation (PARP) inhibitors whereby the process of synthetic lethality can be exploited. In a previous AstraZeneca sponsored Phase II proof of concept study in patients with breast cancer carrying *BRCA* mutations (Study D0810C00008), approximately 60% of cases were *BRCA1* mutations (the other 40% were *BRCA2* mutations) with 55% of tumours overall triple negative in phenotype. In this study, anti-tumour activity was seen in patients with either *BRCA1* or *BRCA2* mutations (<u>Tutt et al 2010</u>).

Given the small size of the *BRCA* subpopulation in breast cancer, information comparing the outcome from this subpopulation with the overall breast cancer population is based on reports from a number of small studies (<u>Robson et al 2004</u>, <u>Rennert et al 2007</u>, <u>Bordeleau et al 2011</u>, <u>Goodwin et al 2012</u>), and firm conclusions cannot be drawn. The overall body of evidence suggests that once baseline prognostic factors (such as hormone receptor and HER2 status) and treatment are taken into account, patients with *BRCA* mutations have a similar outcome to their

sporadic counterparts (<u>Huzarski et al 2013</u>). This is in contrast to patients with *BRCA1/BRCA2*-related ovarian cancer who have an improved survival compared with non-carriers, particularly if they receive platinum-based therapy.

Currently, there are no approved treatments specific for germline *BRCA1/2* mutated breast cancer patients and these patients are treated according to their hormone receptor and HER2 status.

#### 1.1.2 Triple Negative Breast Cancer (TNBC)

TNBC is a particular subset of breast cancer defined by lack or low immunohistochemical expression of ER, PgR and HER2 (IHC 0, 1+ or 2+ /FISH non-amplified) and represents approximately 12-17% of breast cancer overall (Foulkes et al 2010). Although it is a heterogeneous group, patients with TNBC have generally poor prognosis (Metzger-Filho et al 2010). The fundamental clinical characteristic of TNBC is early recurrence with likely early visceral metastases, as well as shorter period from time to recurrence to death as compared with other breast cancer types (Dent et al 2007). Chemotherapy remains the ultimate treatment option for those patients with varied impact on long-term prognosis. No targeted treatment has been developed for TNBC, in contrast to endocrine treatment and anti-HER2 treatments, which have significantly improved the clinical outcomes in ER/PgR positive and HER2 positive breast cancer patients, respectively. The standard clinical practice for early stage TNBC following completion of definitive local and systemic chemotherapy treatment is observation. Therefore, TNBC patients having a poor prognosis and limited treatment options present an unmet need for targeted treatment development.

#### 1.1.3 Adjuvant chemotherapy for TNBC

The majority of patients presenting with early TNBC receive adjuvant chemotherapy. The first randomised Phase III study specifically conducted in early TNBC is the BEATRICE study- an Open Label 2-arm Study to Evaluate the Impact of Adjuvant Bevacizumab on Invasive Disease Free Survival in Triple Negative Breast Cancer (Cameron et al 2013). In this study, 2591 patients with resected early TNBC were randomised to receive adjuvant anthracycline and/or taxane chemotherapy with or without bevacizumab, followed by bevacizumab monotherapy for 12 months. The trial did not meet its primary objective of prolonging invasive disease free survival (IDFS). The 3-year IDFS for both arms of the study was approximately 83%. It was commented that this 3-year IDFS was better than anticipated; however, it should be noted that 63% of patients in the trial were node negative, and ~36% had tumours < 2cm. There are no published robust long-term data for subgroups (e.g. different nodal status or *BRCA* mutated tumours) of TNBC treated with standard of care chemotherapy.

#### 1.1.4 Neoadjuvant chemotherapy for TNBC

It is assumed that approximately a third to half of the patients with TNBC will receive chemotherapy in the neoadjuvant setting. The key prognostic information following neoadjuvant chemotherapy is whether patients have residual disease or have had a pathological complete response (pCR; absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes). Individual patients who achieve pCR following neoadjuvant chemotherapy have significant improvement in both

disease-free survival (hazard ratio (HR) 0.48, 95% CI: 0.37-0.63) and overall survival (HR 0.48, 95% CI: 0.33-0.69) compared with patients with residual invasive disease (Mieog et al 2007). An M.D. Anderson, single institution experience reported 46% pCR rate achieved in a small number of *BRCA1* mutated (n=57) breast cancer patients following anthracycline/taxane neoadjuvant chemotherapy (Arun et al 2011). In TNBC, the prognosis of patients who experience pCR is very similar to that for patients with other breast cancer subtypes with less than 10% developing a distant recurrence at 5 years. However, those patients with TNBC who do not experience pCR have a much poorer prognosis (Liedtke et al 2008, Carey 2011). A recently published meta-analysis of anthracycline and taxane containing neoadjuvant chemotherapy trials showed that of 911 patients with TNBC, 282 patients (31%) experienced a pCR (Von Minckwitz et al 2012). Compared with these patients, patients who did not experience a pCR were at higher risk of earlier recurrence over time (HR 6.02, 95% CI: 3.92-9.25) and at higher risk of earlier death over time (HR 12.41, 95% CI: 5.82-26.49). These results highlight the need to develop further treatment options to improve the prognosis of TNBC patients who do not achieve pCR after neoadjuvant chemotherapy.

#### 1.1.5 ER/PgR positive HER2 negative breast cancer with germline BRCA mutations

While most breast cancers arising in patients with germline *BRCA* mutations are associated histologically with the TNBC phenotype, some - particularly those with underlying germline *BRCA2* mutations - display a non-TNBC phenotype (<u>Honrado et al 2006</u>; <u>Maddavat et al 2012</u>). <u>Atchley et al 2008</u> found positivity for ER /PgR receptor expression in more than 60% of patients with documented germline *BRCA2* mutations and in about 30% of patients with documented *BRCA1* mutations.

Traditionally, these patients have been treated in the same manner as ER/PgR positive patients with either unknown or wildtype *BRCA* status. However, ER/PgR positive, HER2 negative patients with *BRCA2* mutations have been shown to have higher risk of recurrence and death than similar patients without mutations (<u>Tryggvadottir et al 2013</u>), suggesting that the current management of these patients could be suboptimal.

This could be particularly true for high-risk ER/PgR positive, HER2 negative breast cancer patients. Results from NSABP B-38, a trial which employed modern anthracycline and taxane regimens in the adjuvant setting, showed that hormone receptor positive patients with 4 or more positive axillary nodes at surgery had a 3 year DFS of 83%, which is comparable to the 3-year DFS of node negative TNBC (Swain et al 2013).

Similar considerations can be applied to the neoadjuvant setting. In a recently published, FDA co-sponsored meta-analysis looking into the association between the achievement of pCR and long-term clinical benefit, pCR rates in patients with ER and/or PgR positive, HER2 negative tumours were between 8% to 16%, as opposed to 34% in TNBC (Cortazar et al 2014). While all published subgroups in that analysis indicated clinical benefit (longer recurrence-free survival) for those patients achieving a pCR, the associated prognostic value varied *quantitatively* as evidenced by HRs between 0.24 (TNBC patients) and 0.63 (low grade ER and/or PgR positive, HER2 negative tumours with an upper bound of the confidence interval [CI] being slightly above 1.0). A robust association between failure to achieve pCR and event-free survival was demonstrated in patients with ER and/or PgR positive, HER2 negative Grade 3 tumours.

Specifically, the HR for event-free survival in that patient group was found to be almost the same (0.27) as the HR for event-free survival in patients with TNBC (0.24). This demonstrates that for carefully selected, high risk ER and/or PgR positive, HER2 negative patients, failure to achieve pCR can have relatively similar prognostic value as in patients with TNBC who have residual disease after neoadjuvant chemotherapy.

#### 1.1.6 PARP inhibition as a therapeutic strategy target for *BRCA* mutated breast cancer

PARP inhibition is a novel approach to targeting tumours with deficiencies in DNA repair mechanisms. PARP enzymes are essential for repairing DNA single strand breaks (SSBs). Inhibiting PARPs leads to the persistence of SSBs, which are then converted to the more serious DNA double strand breaks (DSBs) during the process of DNA replication. During the process of cell division, DSBs can be efficiently repaired in normal cells by homologous recombination repair. Tumours with homologous recombination deficiencies (HRD), such as ovarian or breast cancers in patients with germline *BRCA1/2* mutations, cannot accurately repair the DNA damage, which may become lethal to cells as it accumulates. In such tumour types, olaparib may offer a potentially efficacious and less toxic cancer treatment compared with currently available chemotherapy regimens.

BRCA1 and BRCA2 defective tumours are intrinsically sensitive to PARP inhibitors, both in tumour models *in vivo* (Rottenberg et al 2008, Hay et al 2009) and in the clinic (Fong et al 2009). The mechanism of action for olaparib results from the trapping of inactive PARP onto the single-strand breaks preventing their repair (Helleday 2011, Murai et al 2012). Persistence of SSBs during DNA replication results in their conversion into the more serious DNA DSBs that would normally be repaired by homologous recombination repair. Olaparib has been shown to inhibit selected tumour cell lines in vitro and in xenograft and primary explant models as well as in genetic BRCA knockout models, either as a stand-alone treatment or in combination with established chemotherapies (data on file at AstraZeneca).

Olaparib is a potent PARP inhibitor (PARP-1, -2 and -3) that is being developed as an oral therapy, both as a monotherapy (including maintenance) and for combination with chemotherapy and other anti-cancer agents.

#### 1.1.7 Pre-clinical experience

The pre-clinical experience is fully described in the current version of the olaparib IB.

#### 1.1.8 Toxicology and safety pharmacology summary

Olaparib has been tested in a standard range of safety pharmacology studies e.g., dog cardiovascular and respiratory function tests, and the rat Irwin test. There were no noticeable effects on the cardiovascular or respiratory parameters in the anaesthetised dog or any behavioural, autonomic or motor effects in the rat at the doses studied.

Rodent and dog toxicology studies have indicated that the primary target organ of toxicity is the bone marrow with recovery seen following withdrawal of olaparib. *Ex vivo* studies have confirmed that olaparib is cytotoxic to human bone marrow cells.

Olaparib was not mutagenic in the Ames test but was clastogenic in the Chinese hamster ovary (CHO) chromosome aberration test *in vitro*. When dosed orally, olaparib also induced micronuclei in the bone marrow of rats. This profile is consistent with the potential for genotoxicity in man.

Reproductive toxicology data indicate that olaparib can have adverse effects on embryofoetal survival and development at dose levels that do not induce significant maternal toxicity.

Further information can be found in the current version of the olaparib IB.

#### 1.1.9 Clinical experience

Clinical experience with olaparib is fully described in the current version of the olaparib IB.

#### 1.1.9.1 Olaparib monotherapy studies in breast cancer patients

#### Study D0819C00003

Olaparib demonstrated a statistically significant improvement in PFS in Study D0819C00003 (OlympiAD), a randomised Phase III study comparing olaparib to chemotherapy of physician's choice (TPC) in the treatment of *gBRCAm* HER2 negative metastatic breast cancer. At 77% maturity, PFS by blinded independent central review was significantly longer in patients treated with olaparib vs. TPC (HR 0.58; 95% CI 0.43-0.80; p=0.0009; 7.0 vs 4.2 months, respectively). Results in the East Asian and White sub-populations were consistent with these findings. PFS2 (time to second progression; investigator-assessed) was also longer in the olaparib arm (HR 0.57; 95% CI 0.40-0.83). Objective response rate was 59.9% and 28.8% in the olaparib and TPC arms, respectively. Final analysis of OS at 64% maturity revealed a median OS of 19.3 months for olaparib vs 17.1 months for TPC (HR 0.90; 95% CI 0.66-1.23) (Robson et al 2017).

#### Study D0810C00002

Study D0810C00002 was a Phase I open-label, dose escalation and cohort expansion study in 98 patients with solid tumours. Patients in the dose-escalation cohort received olaparib at doses ranging from 10 mg daily to 600 mg twice daily (b.i.d.); whereas all patients in the dose-expansion cohort received olaparib at 200 mg twice daily after the MTD was identified as 400 mg b.i.d. The main tumours by type were ovarian (54 [55.1%]), breast, (13 [13.3%]); colon (5 [5.1%]), prostate (4 [4.1%]) and skin cancers (4 [4.1%]). Overall 23 patients were *BRCA* mutation carriers; of these, 19 patients had *BRCA* mutated ovarian, breast, or prostate cancer and were evaluable for response. Forty-seven percent (9/19) of the patients had an objective response as defined by Response Evaluation Criteria in Solid Tumors (RECIST), and 63% (12/19) had stable disease for at least 4 months (Fong et al 2009).

#### Study D0810C00008

Study D0810C00008 was a Phase II proof-of-concept study initiated as an open-label, single-arm, international, multicenter study to assess the efficacy and safety of olaparib given orally b.i.d. in patients with *gBRCA1* and *gBRCA2* mutations and advanced breast cancer. Patients had a median of 3 previous chemotherapy regimens and approximately half of the patients had TNBC. The primary objective was to assess the efficacy of the capsule formulation at 2 different

doses of olaparib in terms of ORR (overall response rate) in patients with advanced breast cancer. Patients received olaparib at a dose of 400 mg b.i.d. or 100 mg b.i.d. continuously in 28-day cycles, for multiple cycles, until no further clinical benefit was apparent or the patient was withdrawn from the study. The cohorts were conducted in sequence, the 400 mg b.i.d. group first (n=27) followed by the 100 mg b.i.d. group (n=27). In the ITT analysis set, the confirmed RECIST ORR overall was 11/27 (41%) at 400 mg b.i.d. and 6/27 (22%) at 100 mg b.i.d. Responses were seen in both gBRCA1 and gBRCA2 carriers. Median time to progression was 5.3 months for the 400 mg b.i.d. group and 3.7 months for the 100 mg b.i.d. group (Tutt et al 2010).

#### Study D0810C00020

Study D0810C00020 was a Phase II open-label, non-randomised study of olaparib in patients with known *gBRCA* or high-grade serous/undifferentiated ovarian cancer and patients with known *gBRCA* or TNBC. All patients received olaparib 400 mg b.i.d. until disease progression or until the investigator believed it was in the best interest of the patient to stop treatment. Tumour response data was analysed in 64 ovarian (*BRCA* or serous ovarian) and 26 breast (*BRCA* or triple negative) cancer patients who received olaparib 400 mg b.i.d. Germline *BRCA* mutations were present in 11 of the 26 breast cancer patients. Median number of prior chemotherapies in the breast cancer group was 3 (range: 1 to 7). Over 70% of the breast cancer patients had received 3 or more previous lines of prior chemotherapy, with a median of 35.3 months from diagnosis to start of treatment with olaparib. None of the breast cancer patients achieved a RECIST response. However, 63% of the patients with *BRCA* mutations had an overall best response of SD lasting 8 weeks or more. The median PFS in this cohort was 3.6 months in this group (Gelmon et al 2011).

#### Study D0810C00042

Study D0810C00042 was a Phase II, open label, non-randomised, non-comparative, multicenter study in patients with advanced cancers who had confirmed germline *BRCA1* and/or *BRCA2* mutations. A total of 62 breast cancer patients were recruited, all of whom received at least 3 prior lines of therapy (with a median of 6 prior regimens). Eight (12.9%) of the breast cancer patients had an OR and the median duration of response was 204 days. At 16 weeks, disease control was observed in 23 (37.1%) patients. The median PFS (progression free survival) was 3.68 months. The median OS was 11.01 months; the survival rate at 6 months was 74.6%, and at 1 year was 44.7% (Kaufman et al 2014).

The details on the pivotal phase II data in ovarian cancer patients as well as olaparib combination with chemotherapy are presented in the Investigator Brochure.

#### 1.2 Research hypothesis

Following completion of definitive local and systemic neoadjuvant or adjuvant chemotherapy treatment, giving olaparib tablet 300 mg b.i.d (twice daily) in the adjuvant setting for up to 12 months in patients with germline *BRCA* mutations and high risk, Stage II-III HER2 negative primary breast cancer has superior efficacy and acceptable tolerability profile as compared with no further treatment. The efficacy in this study will be assessed by the primary analysis of IDFS defined as the time from randomisation to the date of first treatment failure that is loco-regional,

distant recurrence, new invasive cancer or death from any cause. Supportive efficacy analyses include assessment of distant disease free survival and overall survival.

#### 1.3 Rationale for conducting this study

The aim of the proposed phase III study is to obtain a reliable evaluation of whether olaparib monotherapy following completion of definitive local and systemic neoadjuvant or adjuvant chemotherapy is sufficiently safe and provides clinically meaningful benefit in the proposed indication.

The primary endpoint of the trial is IDFS, defined as the time from randomisation to date of first treatment failure that is loco-regional or distant recurrence or new cancer or death from any cause. IDFS is further detailed according to the standardised STEEP system definition (<u>Hudis et al 2007</u>) as one of the following:

- Ipsilateral invasive breast tumour recurrence (IIBTR): invasive breast cancer involving the same breast parenchyma as the original primary.
- Regional invasive breast cancer recurrence: invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast.
- Distant recurrence: metastatic breast cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer.
- Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
- Contralateral invasive breast cancer.
- Second primary non-breast invasive malignancies (i.e. excluding new in situ carcinomas at any site). Second primary non-breast invasive malignancies include hematologic malignancies and MDS. Squamous or basal cell skin cancers will not be counted as primary endpoint events.

Considering the tendency of TNBCs to metastasise to viscera more often than other types of breast cancer, and knowing the generally incurable nature of those with metastases, a secondary endpoint of DDFS will be measured to support the primary endpoint of IDFS and help characterise the secondary endpoint of OS.

In addition to TNBC, the study will also allow patients with positive hormone receptor status as long as they are HER2 negative, who have a germline *BRCA* mutation and fulfil additional criteria for high recurrence risk (see Section 4.1 Inclusion Crit. 3A, 3B, 4b). While events in these patients might not accumulate at exactly the same rate as in *gBRCA*m TNBC, extrapolations from the metastatic setting (Tutt et al 2010) support the expectations that these patients will also benefit from adjuvant olaparib treatment.

In addition, PARP and BRCA function has been linked to estrogen and other hormone receptor transcriptional function (Zhang et al 2013, Schiewer et al 2013), supporting the expectation that

additive/synergistic effects could manifest when combining hormonal treatments with olaparib in hormone receptor positive patients with gBRCAm status. Recent preclinical data by Nardone et al 2015 indicate that olaparib may enhance endocrine therapy efficacy and circumvents resistance; as a consequence, addition of olaparib to hormonal treatment might confer additional treatment benefits in patients with high recurrence risk.

Hence, hormone receptor positive gBRCAm patients will be allowed to receive hormonal treatments at any time during the study. Based on in vitro P450 inhibition and induction data, olaparib would not be expected to alter the PK of standard hormonal therapies used in the adjuvant setting (tamoxifen, aromatase inhibitors with or without ovarian suppression). Based on a preliminary analysis from an ongoing olaparib/hormonal treatment study sponsored by AstraZeneca (Study D081CC00001) there was no indication for clinically relevant drug-drug interaction between olaparib and the anti-hormonal agents tamoxifen, letrozole or anastrozole.

All patients will be followed for local recurrence, distant recurrence (including subsequent sites of recurrence), new cancers and overall survival for a minimum of 10 years, in order to fully describe the long-term impact of adjuvant olaparib therapy.

#### 1.3.1 Rationale for central *BRCA* mutation test at Myriad Genetics, Inc.

The FDA has indicated that the *BRCA1* and *BRCA2* mutation assay will need to be approved as a companion diagnostic in the US.

Myriad Genetics, Inc. has been chosen as a partner in developing a companion diagnostic for *BRCA1* and *BRCA2* testing because it has extensive experience in *BRCA1* and 2 mutation detection. Myriad keeps the most comprehensive database on *BRCA1* and 2 gene mutations and their clinical relevance. Furthermore, Myriad has an established laboratory infrastructure, which supports high volume testing with turnaround times that can meet the needs of a clinical trial.

#### 1.4 Benefit/risk and ethical assessment

As of 20 March 2015, approximately 3862 patients with ovarian, breast, gastric, pancreatic, and a variety of other solid tumours are estimated to have received treatment with olaparib in AstraZeneca-sponsored, investigator-sponsored, and collaborative group studies and a Managed Access Programme. Olaparib has been given as either monotherapy (an estimated 2327 patients) or in combination with other chemotherapy/anticancer agents (an estimated 1535 patients). Many of these combination studies are ongoing. An estimated 1835 patients to date have received the capsule formulation of olaparib, 27 patients have received both the capsule and tablet formulation, and 2000 patients have received the tablet formulation. Approximately 878 patients have received comparator or placebo across the olaparib development programme.

An analysis of monotherapy data across 13 AstraZeneca sponsored monotherapy studies in 1006 patients with ovarian cancer and other non-ovarian solid tumours who have been given olaparib capsules estimated that 16.0% (161/1006) of patients had been exposed to olaparib capsules for  $\geq 12$  months, 8.3% (84/1006) for > 18 months and 4.1% for > 24 months at the time of database closure for the respective studies. Twenty-one patients (2.1%) had received  $\geq 48$  months of olaparib exposure. From the available data to date, there is no evidence of any unexpected toxicity following long-term olaparib (capsule) monotherapy exposure.

In a Phase I study in ovarian cancer patients (Study DO810C00024) the 300 mg b.i.d. monotherapy tablet regimen was considered to have an acceptable tolerability profile relative to the 400 mg b.i.d. capsule and has been determined to be the recommended olaparib monotherapy tablet dose for future studies with olaparib using the tablet formulation. Olaparib as monotherapy at doses up to 400 mg b.i.d. (capsule formulation) and 300 mg b.i.d. (tablet formulation) is generally well tolerated, with most common AEs including nausea, fatigue, vomiting, and anaemia. They were mainly mild-to-moderate (CTCAE Grade  $\leq$  2) in severity.

In addition, in a small number of patients MDS/AML or pneumonitis have been observed and identified as important risks.

#### **Important Potential Risks**

#### Myelodysplastic syndrome/acute myeloid leukaemia

There have been 21 reports of myelodysplastic syndrome (MDS) and/or acute myeloid leukaemia (AML) in patients treated with olaparib as of 20 March 2015; 14 cases in olaparib monotherapy trials and 7 cases in olaparib combination studies with carboplatin and paclitaxel (n=4) or cediranib (n=1), irinotecan and cisplatin (n=2). A total of 3862 patients are estimated to have received olaparib, giving a cumulative incidence of 0.5% for MDS/AML. Two additional reports of MDS have been received from a blinded study (D0816C00002) in which the treatment of the 2 patients (olaparib or placebo) is unknown, and if these patients are considered to have been on olaparib treatment, the estimated incidence would be 0.6%. MDS was also reported for 2 patients who were known to have received placebo or a comparator in the olaparib trial programme (1 patient received placebo in Study D0810C00019 and 1 patient received liposomal doxorubicin in Study D0810C00012). The 21 olaparib-treated patients and two patients on blinded treatment had primary ovarian, peritoneal, fallopian tube cancer (n=20), pancreatic cancer (n=2) or breast cancer (n=1) and 18 of them had germline BRCA1/2 mutations (3 cases BRCA status unknown; 2 cases negative). It has been hypothesised that a deficiency in the expression of BRCA genes may leave patients more vulnerable to the adverse effects of chemotherapy, and therefore, at an increased risk of MDS/AML as a result of cancer treatment (Cole and Strair 2010). Eleven patients had received olaparib for  $\leq 12$  months (5 patients had < 6 months exposure, 6 patients had 6 to 12 months exposure) and the other 12 cases occurred following longer than 12 months olaparib exposure (2 patients following 12-18 months exposure, 2 patients 18-24 months and 8 patients following > 2 years exposure to olaparib).

The median time to onset of t-AML from ovarian cancer diagnosis is reported as approximately 5.5 years (<u>Gupta et al 2007</u>; <u>Vay et al 2011</u>). The overall standardised incidence ratio (8.68 overall) varies over time - 12.07 within 1 to 5 years, 10.81 within 5 to 10 years and 2.30 after 10 years (Morton et al 2013).

Eighteen of the 23 patients died: in 12 of these patients, MDS/AML or myelodysplasia was recorded as either a primary or secondary cause of death. The other 6 deaths were reported as follows: 1 due to cerebral haemorrhage and disseminated intravascular coagulation, 1 due to complication of double umbilical cord blood transplantation and 4 due to disease progression (2 ovarian cancer, 1 breast cancer [patient had a prior history of ovarian cancer treated with platinum-based chemotherapy] and 1 pancreatic cancer). In 5 patients, the event of MDS/AML

is reported as ongoing as of the 20 March 2015. All patients had other potential features that may be contributing factors for the development of MDS/AML. All patients had received previous chemotherapy with DNA damaging agents including platinum, with many patients having extensive previous chemotherapy with multiple treatment regimens over multiple years including carboplatin, taxanes, anthracyclines, other alkylating and DNA damaging agents and radiotherapy.

Since bone marrow is known to be a target organ for olaparib toxicity, increased risk of MDS/AML with long-term exposure to olaparib cannot be excluded. However, there is insufficient data at present to evaluate this relationship. Moreover, while non-clinical data suggest bone marrow progenitor cell populations are reduced temporarily following olaparib treatment, there is no evidence to date linking olaparib treatment to the generation of abnormal bone marrow precursors. Furthermore, all patients who developed MDS/AML had extensive prior chemotherapy and while it is not possible to exclude the contribution of olaparib, it must be considered that there were other potential contributing factors in all cases. Preclinical data also suggest potential benefit with PARP inhibitors in MDS/AML and clinical trials are now underway to assess this effect (Gaymes et al 2008). The risk of developing MDS/AML as a long term toxicity in breast cancer patients with stage I-III disease exposed to standard dose adjuvant chemotherapy including alkylator and anthracycline with or without taxane, is estimated to be around 0.5% varying between 0.37% and 1.16% (Praga et al 2005, Smith et al 2003, Hershman et al 2007, Burnell et al 2010, Aebi et al 2011). Both alkylators and topoisomerase II inhibitors (anthracyclines) have been associated with treatment related MDS/AML. The risk is perceived as low and not outweighing the benefit of adjuvant chemotherapy in breast cancer patients. To ensure robust safety monitoring, patients in this clinical trial will have safety assessments every two weeks during the first month and monthly safety assessments for the first 6 months of treatment followed by 3 monthly assessments until completion of treatment (maximum 12 months treatment). In addition, an Independent Data Monitoring Committee (IDMC) will review the emerging safety data from the trial in an unblinded fashion. Long term safety followup will be implemented in the trial. Clinical guidelines for managing bone marrow toxicity are implemented as part of the safety management plan (Section 5.5.12.4).

#### **Pneumonitis**

As of 20 March 2015, 14 patients out of a total of 3862 patients, estimated to have received olaparib, have reported pneumonitis, giving a cumulative incidence of 0.36% for pneumonitis. Six additional reports of pneumonitis have been received from 4 blinded studies, where the treatment of the patients is unknown (3 either olaparib or placebo; 2 either olaparib + paclitaxel or placebo + paclitaxel and 1 olaparib + abiraterone or placebo + abiraterone). If these patients were considered to have been on olaparib treatment, the estimated cumulative incidence would be 20/3862 (0.52%). Pneumonitis was also reported for 2 patients (1%) of 190 patients that received placebo or comparator in the olaparib trial programme (1 patient on placebo in Study 19 and 1 patient on paclitaxel in Study 39). The patients were treated with olaparib for breast cancer (n=3), ovarian cancer (n=6), non-small cell lung cancer (NSCLC) (n=4), small cell lung cancer (SCLC) (n=1), pancreatic cancer (n=1), gastric cancer (n=3), prostate cancer (n=1) and thymic cancer (n=1). The reports of pneumonitis presented with no consistent clinical pattern and were heavily confounded by a number of pre-disposing factors (including disease under investigation, underlying pulmonary disease, pre-existing medical conditions, smoking history

and/or previous chemotherapy and radiotherapy). The majority of patients had received prior radiotherapy and/or chemotherapy and had other risk factors within the medical histories including pneumonitis, interstitial lung fibrosis, dyspnoea, haemoptysis, chest infection, allergic asthma, pleural effusion, pleural metastases, and smoking. Five patients had current SCLC or NSCLC. An independent review of available chest computed tomography (CT) scans and radiographs associated with the reports of pneumonitis concluded that there appeared to be no clear consistent clinical pattern.

Investigation of any new or worsening pulmonary symptoms has been implemented as part of the safety management plan (Section 5.5.12.5).

#### New Primary Malignancies other than MDS/AML

Overall, the number of reports of new primary malignancies is low, with 24 events (in 22 patients) being reported to 20 March 2015 in 3862 olaparib treated patients (0.57%) and one event (bladder cancer) reported in the placebo arm of the double-blind Study 19. Three additional reports of new primary malignancies have been received from 1 blinded study for the maintenance treatment of ovarian cancer (D0818C00001, tablet formulation), where the treatment of the patients is unknown (either olaparib or placebo). If these patients are considered to have been on olaparib treatment, the estimated cumulative incidence would be 0.65%.

The types of new primary malignancies reported in the 22 patients on olaparib treatment were breast cancer, colon cancer, lung neoplasm malignant, gastric cancer, plasma cell myeloma, basal cell carcinoma, skin cancers, neoplasm skin, squamous cell carcinoma, malignant melanoma, malignant muscle neoplasm, pre-cursor T-lymphocytic lymphoma/leukaemia, tongue cancer and papillary thyroid carcinoma. The 3 patients on blinded treatment reported new primary breast cancer malignancies.

Of the 25 patients (22 on olaparib, 3 on blinded treatment) subsequently diagnosed with a new primary malignancy, the majority were reported whilst receiving study treatment (21 patients). In 4 patients the event was reported after olaparib discontinuation (within 60 days after olaparib discontinuation in 2 patients, and more than 240 days after olaparib discontinuation in 2 patients).

The duration of treatment for the 25 patients was

- <6 months for 5 patients
- 6 to 12 months for 8 patients
- 12 to 18 months for 2 patients
- 18 to 24 months for 3 patients
- >2 years for 7 patients.

The type of new primary cancers reported were generally in line with secondary cancers observed in ovarian and breast cancer populations reported in the literature (<u>Bergfeldt et al 1995</u>,

<u>Fowble et al 2001</u>, <u>Wesolowski et al 2007</u>), or were cancers such as skin cancer, known to be the most common cancer in the general population and associated with high cure rates.

Ovarian cancer patients have been reported to have an increased risk of developing second primary malignancies. Patients with germline BRCA mutations are at risk of developing other primary cancers notably breast cancer. Ginsburg et al 2010 reported higher rates of skin cancers in patients with BRCA1 (1.6%) and BRCA2 (3.0%) mutations.

There were other contributing factors/potential alternative explanations for the development of the new primary malignancy in all 22 olaparib treated patients and the 3 on blinded treatment. All patients had previously received various chemotherapy agents including multiple cycles of DNA damaging platinum containing chemotherapies, taxanes, anthracyclines and other alkylating and DNA damaging agents. Four patients were reported to have had prior radiotherapy. Twenty-two patients had a documented breast cancer gene mutation (*BRCA* 1 or 2). Seven of the 25 patients had previous medical histories of cancer (ovarian, cervix, breast, peritoneal) and 3 patients with skin cancers either had previous basal cell carcinoma reported or skin lesions evident prior to study treatment.

There is insufficient evidence for an association between olaparib treatment and the development of new primary malignancies in the clinical trial programme to date. The risk is perceived as low and not outweighing the benefit of adjuvant chemotherapy in breast cancer patients. An IDMC will review the emerging data from the trial in an unblinded fashion.

#### **Potential benefit**

A Marketing Authorisation Application was approved in EU/EEA on 16 December 2014 for the indication 'LYNPARZA monotherapy for the maintenance treatment of adult patients with platinum-sensitive relapsed BRCA-mutated (germline and/or somatic) high grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in response (complete response or partial response) to platinum-based chemotherapy.'

A New Drug Application was approved in the US on 19 December 2014 for the indication 'LYNPARZA monotherapy in patients with deleterious or suspected deleterious germline BRCA mutated (as detected by an FDA-approved test) advanced ovarian cancer who have been treated with three or more prior lines of chemotherapy.'

Olaparib tablet formulation was approved in January 2018 for patients with deleterious or suspected deleterious *gBRCAm*, HER2-negative metastatic breast cancer who have previously been treated with chemotherapy in the neoadjuvant, adjuvant or metastatic setting. Patients with hormone receptor-positive breast cancer should have been treated with a prior endocrine therapy or be considered inappropriate for endocrine treatment.

Phase II clinical studies have investigated the effect of olaparib either as monotherapy or in combination with other chemotherapy agents in cancer patients. In patients carrying germline BRCA mutations, monotherapy studies in patients with heavily pre-treated breast cancer have reported an ORR of up to 41%.

In ovarian cancer patients, the pivotal phase II study D0810C00019, a double-blind, randomised study assessed the efficacy of olaparib 400 mg b.i.d. capsules as a maintenance treatment
following platinum-based chemotherapy in patients with platinum sensitive relapsed high grade serous ovarian cancer. The PFS following olaparib maintenance therapy was significantly longer compared with the placebo group (HR 0.35; 95% CI: 0.25, 0.49; p<0.00001) in the overall population. In the subgroup of patients with *BRCA* mutant ovarian cancer, the effect was even greater with a PFS HR of 0.18 (95% CI: 0.11, 0.31; p<0.00001; median 11.2 versus 4.3 months). An interim analysis of OS was performed at 58% maturity. In the overall population, the analysis demonstrated a non-statistically significant numerical advantage for olaparib-treated patients (OS HR 0.88; 95% CI 0.64-1.21; p=0.43808) and there was again a greater effect in the *BRCA*-mutated subgroup: the OS HR was 0.74 (95% CI 0.46 to 1.19; p=0.20813) with a numerical advantage in median OS observed with olaparib (median 34.9 months versus 31.9 months with placebo). Among the 62 placebo-treated patients with *BRCA* mutations, 14 switched to a PARP inhibitor post progression.

Based on these results and data from the full clinical program to date, it is anticipated that in the adjuvant setting, olaparib will have a positive benefit risk profile for the treatment of the small well-defined population of high-risk HER2 negative primary breast cancer patients with *BRCA* mutations.

#### 2. STUDY OBJECTIVES

# 2.1 Primary objective

The primary objective is to assess the effect of adjuvant treatment with olaparib on Invasive Disease Free Survival (IDFS).

# 2.2 Secondary objectives

The secondary objectives of this study are:

- 1. To assess the effect of adjuvant treatment with olaparib on overall survival (OS)
- 2. To assess the effect of adjuvant treatment with olaparib on Distant Disease Free Survival (DDFS)
- 3. To assess the effect of adjuvant treatment with olaparib on the incidence of new primary contralateral breast cancers (invasive and non-invasive), new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer
- 4. To assess the effect of olaparib on patient reported outcomes using the FACIT-Fatigue and EORTC QLQ-C30 questionnaires
- 5. To assess the efficacy of olaparib in patients identified as having a deleterious or suspected deleterious variant in either of the *BRCA* genes using variants identified with current and future *BRCA* mutation assays (gene sequencing and large rearrangement analysis)
- 6. To determine the exposure to olaparib (in plasma) in patients receiving olaparib as adjuvant therapy

# 2.3 Safety objective

To assess the safety and tolerability of adjuvant treatment with olaparib

| Redacted | Redacted |
|----------|----------|
| Redacted | |
| Reda | Redacted |
| Reda | Redacted |
| _ | |
| _ | |

# 3. STUDY PLAN AND PROCEDURES

This Clinical Study Protocol has been subject to a peer review according to AstraZeneca standard procedures.

# 3.1 Overall study design, flow chart and study schedules

This is a randomised, double-blind placebo controlled multicentre, phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy.

Randomised patients will receive study treatment for up to a maximum of 12 months. All patients will have safety assessments every 2 weeks during the first month, every 4 weeks for the following 5 months (up to week 24) and 3 monthly for the remaining 6 months of study treatment, plus 30 days after its discontinuation. Efficacy assessments (medical history and physical examination) will be performed on a 3 monthly basis during the first 2 years following end of study treatment, followed by 6 monthly assessments for years 3, 4 and 5 and annually thereafter. Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory before enrolment (within 12 months prior to Screening PART 1) and during study participation (starting at week 24 and yearly thereafter) for patients with any remaining intact breast tissue. The preferred tests are mammogram or magnetic resonance imaging (MRI; MRI preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion. Evidence of disease recurrence or new primary cancer will require histopathological and/or radiological confirmation.

Patients who develop loco-regional recurrence should have cytological/histological confirmation. Loco-regional recurrence should be treated with curative intent when possible. Appropriate imaging (CT, MRI bone and/or PET scan) of the chest/abdomen/pelvis or any other area as clinically indicated (MRI preferred to examine CNS (central nervous system) if new neurological symptoms occur) should be performed at the time of local recurrence to exclude further spread of the disease.

Distant recurrence should be diagnosed by radiological/imaging examination and every attempt should be made for histopathological confirmation when metastatic lesion is accessible for biopsy.

If the patient meets the IDFS endpoint due to a breast cancer related distant relapse, the patient will enter the survival follow-up phase of the trial, with annual assessments from the date of distant relapse, which will continue until 10 years after the last patient is randomised. No clinic visits will be required during the survival follow-up phase; information may be collected via telephone, medical records or death registries. During the survival follow-up phase, in addition to vital status, the following information will be collected (if available): specific cancer therapies (only first line treatment for first breast cancer recurrence and any subsequent regimens

containing PARP inhibitors or platinum received by the patient at any time), sites of metastases and any other new cancer.

If the IDFS endpoint is met due to events other than distant relapse, the patient will continue the efficacy assessment visit study schedule until breast cancer related distant relapse occurs, or approximately 10 years following their randomisation into the study, whichever occurs first. They will then enter the survival follow-up phase of the trial.

See <u>Section 5.8.1</u> for guidelines on study visits for any patient discontinuing prior to completing 52 weeks of study treatment.

Figure 1 Study Flow Chart

ICF for patients with unknown *BRCA* status to undergo central *BRCA* testing during, or prior to, neoadjuvant/adjuvant chemotherapy



Patients will continue to be followed clinically on a 3 monthly basis during the first 2 years, followed by 6 monthly assessments for the 3rd, 4th and 5th year, and annually thereafter

Yearly breast imaging (mammogram **and/or** MRI) (ipsilateral and/or contralateral) for 10 years\*

\*The study will end 10 years after the last patient has been randomised

# Figure 2 Screening Plan

# Screening PART 1 – Patients with Unknown gBRCA Mutation Status:

• Only those patients who **do not** know their gBRCA mutation status prior to entry in to the study These patients will undergo screening assessments as described for PART 1 in <u>Table 1</u>. Screening PART 1 is conducted to determine if the patient is considered **eligible to undergo the** BRCA **status blood test**. Once PART 1 has been successfully completed and patients have had a BRCA test, these patients will continue to PART 2 and have all procedures performed as described for PART 2 (see <u>Table 1</u>)

# Screening – PART 2 – ALL Patients (Patients with Known gBRCA Mutation Status):

- Those patients who already know their gBRCA mutation status **and** have a deleterious or suspected deleterious mutation to undergo screening assessments as described for PART 2 (see <u>Table 1</u>)
- Those patients originally with unknown gBRCA status who have completed screening PART 1 and now have a confirmed deleterious or suspected deleterious mutation should undergo screening assessments as described for PART 2 (see <u>Table 1</u>)

Table 1 Study Schedule - Screening (PART 1 and PART 2)

| Day | Any time prior, during or after neoadjuvant/adjuvant chemotherapy or radiotherapy PART 1 a (ONLY Patients requiring a gBRCA status Myriad test before randomisation) | -28 to 0 days PART 2 (Patients with confirmed gBRCA status by Myriad or if BRCA status is known prior to study entry j) |
|---|---|---|
| Informed consent | X b,c | Хj |
| Demographics (date of birth) | X | X |
| Medical and surgical history d | | X |
| Prior cancer therapies including radiotherapy | | X |
| Inclusion/exclusion criteria | X (all ** criteria) | X |
| ECOG Performance Status | | X |
| Physical examination | | X |
| Vital signs | | X |
| ECG f | | Хg |
| Haematology / clinical chemistry/Coagulation 0 | | X |
| Urinalysis h | | X |
| Pregnancy test i | | X |
| EORTC QLQ-C30 n | | X |
| FACIT-Fatigue n | | X |
| Blood sample for determination of <i>BRCA</i> status via Myriad | X | Хе |
| Blood sample for assessment of current and future <i>BRCA</i> mutation assay(s) <b>c</b> | X | Хе |
| Concomitant medications | | X |
| Archival tumour sample (FFPE) (mandatory) k | | X |
| Surgical tumour sample (FFPE) (post neoadjuvant chemotherapy (mandatory)) k | | X |

Table 1 Study Schedule – Screening (PART 1 and PART 2)

| Day | Any time prior, during or after neoadjuvant/adjuvant chemotherapy or radiotherapy PART 1 a (ONLY Patients requiring a gBRCA status Myriad test before randomisation) | -28 to 0 days PART 2 (Patients with confirmed gBRCA status by Myriad or if BRCA status is known prior to study entry j) |
|---|---|---|
| Radiological assessment to exclude metastatic breast cancer (where applicable) l | | X |
| Family history of cancer | | X |
| Serious Adverse Events m | X (only SAEs due to study procedures) | X (SAEs only) |

- a The time period is to allow those patients that require a Myriad gBRCA sample to have the test taken and the results returned prior to randomisation.
- b It is recommended that patients that require the Myriad gBRCA sample testing are to be consented for BRCA testing and participation in the trial prior or during neoadjuvant/adjuvant chemotherapy prior to entering the study.
- c Any patient who consents to study related Myriad gBRCA status testing, must also have a blood sample taken at the same time for the purpose of developing and validating a future mutation assay.
- d Include history of blood transfusion within previous 120 days from start of study treatment and the reasons e.g. bleeding. Additionally CPS+EG score components should be collected (Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS)) for the non-pCR patients who received prior neoadjuvant chemotherapy. Instructions on how to calculate the CPS&EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix H.
- e Samples to be taken in screening PART 2 only for patients with known gBRCA mutation who have not completed PART 1.
- f ECG recordings should be performed once the patient has been in the supine position for at least 5 minutes.
- g ECG assessments to be completed within 28 days before randomisation.
- h Urinalysis (dipstick) should be performed at screening. After screening, urinalysis will only be required if clinically indicated.
- i Women who are not postmenopausal or have not undergone hysterectomy must have a negative urine or serum pregnancy test within 28 days prior to randomisation and a confirmatory test on Day 1 before starting study treatment. If the results are positive the patient is ineligible.
- j Patients for whom their gBRCA status is already known, should be consented to the study within 28 days prior to randomisation.
- k Mandatory for all randomised patients i.e. for adjuvant patients this refers to the surgical specimen; for neoadjuvant patients, both the pre-treatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required. Samples will only be sent to the study bio-repository once the patient has been randomised.
- Patients considered at high risk of having disseminated disease (i.e. those with locally advanced disease, clinical N2-3 or pathological N1-3 with the exception of pN1a in adjuvant patients are expected to have a CT/MRI scan of the Thorax/Abdomen/Pelvis or any other area as clinically indicated and a bone scan <u>or</u> a CT scan with bone windows at any point between diagnosis of the current breast cancer and randomisation to rule

out metastatic breast cancer. (Note PET/CT scan may be used as an alternative imaging technique and precludes the need for bone scan). Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory before enrolment (within 12 months prior to Screening PART 1) for patients with any remaining intact breast tissue. The preferred tests are mammogram or MRI (MRI preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion.

To rule out metastatic breast cancer, patients with screening ALT/AST or ALP above institutional upper limit of normal should have liver ultrasound, CT or MRI at any time point between diagnosis of current breast cancer and randomisation. Screening bone scan is required if ALP and/or corrected calcium level are above the institutional upper limit. (Note PET/CT scan may be used as an alternative imaging technique).

- m Serious adverse events must be captured from time of consent. In Screening PART 1 of the study only SAEs related to a study procedure will be collected. In Screening PART 2 all SAEs will be collected.
- n EORTC QLQ-C30 + FACIT-Fatigue will be collected prior to randomisation once eligibility is confirmed.
- o Coagulation analysis only required at baseline.

| (Year 1 |
|----------------|
| On treatment ( |
| Jule – ( |
| / Schedul |
| Study Sche |

| | | | | ( , | | | |
|---|---|---|---|---|---|---|---|
| Visit Number | 7 | က | 4 | 5-9 | 10-11 | Premature study | Follow-up 30 days |
| | | | | (Every 4 weeks) | (Every 3 months (14 weeks)) | treatment<br>discontinuation g | after last dose of study medication (all patients) |
| Week | 0 | 2 | 4 | 8, 12, 16, 20, 24 | 38, 52 | | |
| Day | - | 15 | 29 | | | | |
| Visit Window | | <del>+</del> 3d | ∓3d | ±1 week | ±2 week | +2 week | +2 week |
| Serum or urine pregnancy test for women of childbearing potential a | X | | × | X | X | | X |
| ECOG performance status | q X | | | | | | |
| Vital signs | Хр | | X | X (weeks 12 and 24 only) | X | X | X |
| Haematology / clinical<br>chemistry <b>c</b> | X b,c | X | X | X | X | X | X |
| Recurrent/new cancers assessment (includes physical exam d, clinical signs and symptoms) | X | | | X (weeks 12 and 24 only) | X | X | X |
| Mammogram and/or breast<br>MRI (ipsilateral and/or<br>contralateral) (MRI preferred<br>for patients younger than<br>50 years) e | | | | X (week 24 only) | | | |
| Adverse Events | X | X | X | X | X | X | X |

| Year 1 |
|---------------|
| $\overline{}$ |
| treatment |
| $\frac{1}{2}$ |
| 0 |
| Ξ |
| Ę |
| ĕ |
| _ |
| ٢ |
| 7 |
| Ħ |
| S |
| •1 |
| (1 |

| Table 2 Study Schedule – On treatment (Year 1) | le – 0 | n trea | tment | (rear 1) | | | |
|---|---|---|---|---|---|---|---|
| Visit Number | 7 | e | 4 | 8-9 | 10-11 | Premature study | Follow-up 30 days |
| | | | | (Every 4 weeks) | (Every 3 months (14 weeks)) | treatment<br>discontinuation g | after last dose of<br>study medication<br>(all patients) |
| Week | 0 | 2 | 4 | 8, 12, 16, 20, 24 | 38, 52 | | |
| Day | 1 | 15 | 29 | | | | |
| Visit Window | | ±3d | ±3d | ±1 week | ±2 week | +2 week | +2 week |
| Concomitant medications including blood transfusions | × | × | × | X | X | X | X |
| Demographics j | X | | | | | | |
| EORTC QLQ-C30 | | | | X (week 24 only) | X (week 52 only) | | |
| FACIT-Fatigue | | | | X (week 24 only) | X (week 52 only) | | |
| Biomarker Blood 2 samples (mandatory) | Xi | | | | | | X |
| PGx Blood sample (optional) | × | | | | | | |
| Blood sample for PK analysis (optional; after signing PK Informed consent) (subset of patients) h | | | × | | | | |
| Blood biomarker samples at disease recurrence (Mandatory) | × | × | × | X | X | X | X |
| Tumour biopsy at disease recurrence (Optional) <b>k</b> | × | X | X | X | X | X | X |
| Olaparib dispensed/returned f | X | | X | X | X | X | |

If assessed within 7 days before randomisation, it does not need to be repeated on Day 1 of study treatment unless investigator believes that it is likely to have changed significantly. 9

Safety blood samples do not need to be repeated on Day 1 of study treatment if they have been assessed within 7 days before randomisation and which must Safety bloods samples are to be collected every 2 weeks during the first 4 weeks, then every 4 weeks until week 24 and then at weeks 38 and 52 of study have been done at least 3 weeks after the last dose of chemotherapy, unless the investigator believes that they are likely to have changed significantly.

Physical examination both local and general should be performed at day 1 and then at weeks 12, 24 and 38 and 52 post randomisation until study treatment is discontinued (data is not required to be captured on an eCRF, however any significant changes from baseline must be reported as an AE) 7

tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and radiological Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory during study participation (starting at week 24 and yearly thereafter) for patients with any remaining intact breast tissue. The preferred tests are mammogram or MRI (MRI preferred for patients below exams at investigator's discretion.

Sufficient study treatment should be dispensed for at least each treatment period plus overage, however additional treatment can be dispensed to patients to last longer in accordance with local practice.

met due to breast cancer related distant relapse, the patients enters the survival follow-up phase and is assessed annually from the date of distant relapse and inhibitors or platinum received by the patient at any time), sites of metastases and any other new cancers. If a recurrent/new cancer assessment is scheduled until 10 years after the last patient is randomised. In case the IDFS endpoint is met due to other events, the patient will continue the study schedule until a collected (if available): specific cancer therapies (only first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP breast cancer related distant relapse occurs or approximately 10 years following their randomisation into the study, whichever occurs first. They will then regimens containing PARP inhibitors or platinum received by the patient at any time) should also be recorded on the eCRF. In case the IDFS endpoint is followed by the 30-day follow-up visit and site staff completes relevant CRF pages as required. In case of premature treatment discontinuation, only the enter the survival follow-up phase of the trial. During the annual survival follow-up phase, in addition to vital status, the following information will be visits where efficacy assessments are scheduled should be performed i.e. week 12, 24, 38, 52 (as applicable) in Year 1 and all visits in Year 2 onwards. discontinuation, the reasons, and details of the following specific cancer therapies (first line treatment for breast cancer recurrence and any subsequent therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse. The date of If a patient discontinues prior to completing 52 weeks of study treatment, the patient should have the study treatment discontinuation visit performed Collection of vital signs, AEs, haematology/clinical chemistry results, and concomitant medications is no longer required. Information on endocrine within 4 weeks of the study treatment discontinuation visit, it can be performed at the 30 day follow-up visit (for more details see Section 5.8.1) ba

PK sampling (optional) to be performed in a subset of patients. Sampling times: pre-dose (before morning dose) plus one sample in each of the following sampling windows: 0 to 0.5 h post dose, > 0.5 to 1.5 h post dose, 3 to 6 h post dose and > 6 to 12 h post dose (before evening dose) preferably on visit 4, day 29. Nevertheless, the samples can also be taken at a later treatment visit, provided that PK consent was obtained beforehand (for details see Section Ч

Blood samples (plasma and serum) for biomarker analysis should be collected on Day 1 prior to first dose of study treatment.

j Race and ethnicity to be collected unless not allowed by local regulation.

**NSABP B-55/BIG 6-13** NCI Version Date: 05-06-2021

Table 3 Study Schedule - Follow-up Visits (Year 2 onwards)

| Visit Number | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | Survival<br>Follow-up<br>(Every 12<br>months) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Year | | 2 | | | 3 | | 4 | | 5 | | 9 | 7 | 8 | 6 | 10 | 11+ |
| Month | 15 | 18 | 21 | 24 | 30 | 36 | 42 | 48 | 54 | 09 | 99 | 78 | 06 | 102 | 114 | 126, 138,<br>etc. |
| Visit Window | | ±1 m | month | | | | ±2 months | nths | | | | # | ±3 months | ths | | ±3 months |
| Recurrent/new cancers assessment (includes physical exam, clinical signs and symptoms) | X | X | X | × | × | × | X | X | X | X | X | X | X | X | X | |
| Mammogram and/or breast MRI (ipsilateral and/or contralateral) (MRI preferred for patients younger than 50 years) a | | × | | | × | | × | | X | | × | × | × | X | X | |
| Subsequent cancer therapy <b>b</b> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | рХ |
| Overall survival assessment | | | | | | | | | | | | | | | | рΧ |
| EORTC QLQ-C30 | | X | | X | | | | | | | | | | | | |
| FACIT-Fatigue | | X | | X | | | | | | | | | | | | |
| Blood biomarker samples at disease recurrence (Mandatory) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Tumour sample at disease recurrence (Optional) c | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| SAEe | X | × | × | × | × | × | × | X | × | X | X | X | X | X | X | X |

- ime need to be recorded. Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to First line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any breast cancer related distant relapse. 9
- The provision of tumour tissue is encouraged only if clinically appropriate and not considered detrimental to patient care and patient agreed to the optional tumour biopsy in the consent form.
  - During the annual survival follow-up phase, information (where available) on further subsequent cancer therapies (see footnote b), sites of metastases and any other new cancers will be collected in addition to vital status.
- 30-day follow-up period should be reported as a SAE, regardless of investigator's assessment of causality, knowledge of the treatment arm, and irrespective of the timing of the event in relation to study therapy. Non-melanoma invasive skin cancers and all cases of carcinoma in situ need to be reported as a nonfollowed to resolution unless the event is considered by the investigator to be unlikely to resolve, or the patient is lost to follow-up or in survival follow-up serious AE unless at least one of the seriousness criteria is met which then requires reporting as a SAE, see Section 6.4.6. If a patient develops MDS/AML If an investigator learns of any SAEs, including death, at any time after a patient has completed the 30 days post treatment follow-up period, and he/she questionnaire will be sent to any investigators reporting MDS/AML or new primary malignancies as an aid to provide detailed information on the case. reporting procedures for this study. Any cases of MDS/AML, any new second primary malignancies or diagnoses of pneumonitis occurring after the 'ull diagnostic details and classification should be provided e.g. bone marrow and cytogenetic analysis reports, see Sections 5.5.12.4 and 6.4.11.5. A considers there is a reasonable possibility that the event is causally related to the study treatment, the investigator should report it according to SAE All ongoing AEs/SAEs and any new AEs/SAEs identified during the 30 calendar days follow-up period after last dose of study medication must be

# 3.2 Rationale for study design, doses and control groups

# 3.2.1 Rationale for study design

In this placebo-controlled, double-blinded adjuvant study, TNBC patients and ER and/or PgR positive HER2 negative patients with germline *BRCA* mutations at high risk of recurrence will be randomised to receive monotherapy olaparib 300 mg tablet b.i.d. (twice daily) or corresponding placebo for a maximum of 12 months following completion of their definitive loco-regional treatment and chemotherapy in the adjuvant or neoadjuvant setting.

The rationale for allowing patients with ER and/or PgR positive HER2 negative breast cancer who carry a *gBRCA*m (including gene rearrangements) is provided in <u>Section 1.3</u>.

The use of a placebo comparator to olaparib is considered acceptable in order to objectively test the hypothesis of improved efficacy with the addition of olaparib for up to 12 months as compared to no further therapy (i.e. placebo) in patients with TNBC and endocrine therapy alone in patients with ER and/or PgR positive cancer. By blinding patients and investigators, using placebo control and assessing patients for the disease recurrence at pre-defined intervals, the risk of bias that could affect the interpretation of the IDFS endpoint should be minimised. In line with international clinical guidelines evidence of disease recurrence will be assessed during the regular follow-ups (3 monthly during the first 2 years, 6 monthly during the 3rd, 4th and 5th year and annually afterwards) by medical history, physical examination and mammogram and/or breast MRI (MRI preferred for patients younger than 50 years) (ipsilateral and/or contralateral), unless clinical signs and symptoms require further investigation (Khatcheressian et al 2012). In addition safety follow-ups are implemented during the 12-month study treatment period and 30 days after its discontinuation.

It should be noted that the safety and efficacy of olaparib has been demonstrated in the clinical program using the capsule formulation (400 mg - 8 capsules - twice daily); however, an improved tablet formulation (2 tablets twice daily) has been developed and will be used in this study. The tablet dose of olaparib that will be investigated is 300 mg b.i.d. (twice daily) which is considered similar to the capsule 400 mg b.i.d. (twice daily) dose. This tablet dose has been chosen based on data from Study D0810C00024. Since it has been shown that the capsule and tablet formulations are not bioequivalent, a formulation switch based on bioequivalence has not been possible. The tablet dose of 300 mg b.i.d. is considered to have similar efficacy in terms of tumour shrinkage in ovarian cancer patients with BRCA mutations to the 400 mg b.i.d. capsule. The 300 mg b.i.d. tablet dose matches or exceeds the exposure of the 400 mg capsule in terms of AUC,  $C_{maxss}$ , and  $C_{minss}$ . The tolerability profile of the 300 mg b.i.d. tablet dose in Study D0810C00024 was considered similar to the 400 mg b.i.d. capsule formulation. The most common AEs were consistent with the known safety profile of olaparib, namely low grade nausea, vomiting, fatigue, and anaemia. Further information is provided in the olaparib Investigator's Brochure.

# 3.2.2 Rationale for patient reported outcomes

The patient population for this study will have had intensive treatments with chemotherapy (neoadjuvant or adjuvant), surgery, and possibly radiation therapy prior to entry and randomisation on this study. Prior research by the NSABP and other investigators has

NCI Version Date: 05-06-2021 55(177) NSABP B-55/BIG 6-13

demonstrated physical disruption and many symptoms at the end of primary treatment (<u>Ganz et al 2011B</u>, <u>Ganz et al 2004</u>). Research has shown that it may take a year or more for the physical and emotional recovery and that symptoms may persist well beyond improvements in health related quality of life (HRQoL) (<u>Ganz et al 2011A</u>, <u>Ganz et al 1998A</u>, <u>Ganz et al 1998B</u>, <u>Ganz et al 2002</u>, <u>Bower et al 2000</u>, <u>Bower et al 2006</u>). Thus, in any studies that are designed to capture patient-reported outcomes (PROs) of treatment, consideration should be given to assessment of both HRQoL and symptoms.

In this trial of olaparib versus placebo, there is an important opportunity to determine whether or not the use of olaparib delays or retards recovery after primary breast cancer treatment, and if so, what aspects of symptoms and HRQoL are impaired. Gelmon et al 2011 reported on a Phase II open label study of olaparib in breast and ovarian cancer patients, in which fatigue was the most common reported toxicity (50-70% of patients) followed by nausea (62-66%), vomiting (35-39%), and decreased appetite (27-36%). In a Phase II study in patients with *BRCA1* or *BRCA2* mutations and advanced breast cancer, fatigue was the most significant toxicity (41% grade 1-2, and 15% grade 3-4) in the cohort given 400 mg twice daily (Tutt et al 2010). These trials did not use PROs, and since they were conducted in patients with advanced disease, there is uncertainty about how much fatigue patients will have in the B-55/6-13 trial. However, since this is the most frequent side effect of olaparib, it is our primary outcome in this placebo-controlled comparison.

The FACIT-Fatigue scale will be used to measure treatment related fatigue. The FACIT-Fatigue measure that is being used in this study is well-established and available in multiple languages.

A standard measure of health-related cancer specific HRQoL, the EORTC QLQ-C30, will be used in this study to track recovery in key domains of HRQoL in the year after initial treatment, and to measure symptoms, with a heightened focus on fatigue and GI symptoms (nausea, vomiting, diarrhea), as these symptoms have been reported with olaparib. The GI symptoms items from the EORTC QLQ-C30 will be used to assess their severity, with the focus on assessments during the treatment period, and in the year following the end of treatment. These self-report instruments have been selected for this study due to the need for reliable and valid translations in multiple languages, given the international scope of this trial and the need to include a large number of participants.

Refer to Section 12.2.3 for patient reported outcomes hypotheses and objectives.

# 3.2.3 Study Population

Approximately 1800 patients with germline *BRCA* mutations (*gBRCA*m) and HER2 negative breast cancer who are at high risk of recurrence will be randomised into the trial.

All patients recruited in the study will be selected based on the following 3 principles:

• **Genetic selection**: Documented germline mutation in *BRCA1* or *BRCA2* that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function). Patients with germline *BRCA1* and/or germline *BRCA2* mutations that are considered to be non-detrimental (e.g. "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favour polymorphism" or "benign

NCI Version Date: 05-06-2021 56(177) NSABP B-55/BIG 6-13

polymorphism," etc) will not be eligible for the study. In terms of *BRCA* mutation status, the following scenarios are considered:

- Status known: for patients already known to have a gBRCA loss of function mutation (known as deleterious or suspected deleterious) the exact sequence variant must be recorded on the eCRF and a copy of the genetic diagnosis must be available at site. These patients may be randomised into the study based on the known status; however, re-confirmation of the loss of function mutation from a blood sample will be undertaken soon after randomisation by Myriad Genetics, Inc.
- Status unknown: The gBRCA mutation status must be determined by Myriad Genetics, Inc. prior to randomisation as a loss of function mutation i.e. a known deleterious or suspected deleterious mutation
- **Phenotypic tumour selection**: All patients must have either TNBC or ER and/or PgR positive HER2 negative breast cancer as defined in the eligibility criteria section.
- **Prognostic factor selection**: Patients will be selected based on high risk of recurrence regardless of whether they received their chemotherapy in the adjuvant or neoadjuvant setting. High risk of recurrence will be defined as follows:
  - 1. For patients who underwent initial surgery and received adjuvant chemotherapy
    - TNBC patients must have been axillary node-positive (≥pN1, any tumour size) or axillary node negative (pN0) with invasive primary tumour pathological size > 2 cm (≥pT2)
    - ER and/or PgR positive/HER 2 negative patients must have had ≥4 pathologically confirmed positive lymph nodes
  - 2. For patients who underwent neoadjuvant chemotherapy followed by surgery
    - TNBC patients must have residual invasive breast cancer in the breast and/or resected lymph nodes (non pCR)
    - ER and/or PgR positive/HER 2 negative patients must have residual invasive cancer in the breast and/or the resected lymph nodes (non pCR) AND a CPS&EG score ≥3. Instructions on how to calculate the CPS&EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix H.

NCI Version Date: 05-06-2021 57(177) NSABP B-55/BIG 6-13

#### 4. PATIENT SELECTION CRITERIA

Investigator(s) should keep a patient screening log of patients who entered pre-study screening.

Each patient should meet all of the inclusion criteria and none of the exclusion criteria for this study. Under no circumstances can there be exceptions to this rule.

Criteria relevant to Part 1 BRCA screening (Table 1) are marked with (\*\*) double asterisk

#### 4.1 Inclusion criteria

For inclusion in the study patients should fulfil the following criteria:

- 1. \*\*Provision of informed consent prior to any study specific procedures
- 2. \*\*Female or male patients must be ≥18 years of age
- 3A. For patients who underwent initial surgery and received adjuvant chemotherapy
  - TNBC patients must have been axillary node-positive (≥pN1, any tumour size) or axillary node-negative (pN0) with invasive primary tumour pathological size
     2 cm (≥pT2)
  - ER and/or PgR positive/HER 2 negative patients must have had ≥4 pathologically confirmed positive lymph nodes
- 3B. For patients who underwent neoadjuvant chemotherapy followed by surgery
  - TNBC patients must have residual invasive breast cancer in the breast and/or resected lymph nodes (non-pCR)
  - ER and/or PgR positive/HER2 negative patients must have residual invasive cancer in the breast and/or the resected lymph nodes (non-pCR) AND a CPS&EG score ≥3. Instructions on how to calculate the CPS&EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix H.
- 4. \*\*Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast that is one of the two following phenotypes:
  - a) TNBC defined as:
    - ER and PgR negative defined as IHC nuclear staining <1%.

**AND** 

- HER2 negative (not eligible for anti-HER2 therapy) defined as:
  - o IHC 0, 1+ without ISH **OR**

NCI Version Date: 05-06-2021 58(177) NSABP B-55/BIG 6-13

- o IHC 2+ and ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells **OR**
- o ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells (without IHC)
- b) ER and/or PgR positive, HER2 negative breast cancer defined as:
  - ER and/or PgR positive defined as IHC nuclear staining  $\geq 1\%$ .

#### **AND**

- HER2 negative (not eligible for anti-HER2 therapy) defined as:
  - o IHC 0, 1+ without ISH **OR**
  - o IHC 2+ and ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells **OR**
  - O ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells (without IHC)

Patients with multifocal or multicentric invasive disease are eligible as long as all the lesions for which HER2 characterization is available are HER2 negative.

Patients with synchronous bilateral invasive disease are eligible as long as all the lesions assessed for HER2 on both sides are negative.

In both the above cases, the lesion considered at highest risk for recurrence based on the investigator's discretion will be used for eligibility determination.

- 5. Documented germline mutation in *BRCA1* or *BRCA2* that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function). Local *gBRCA* testing results, if available, will be used for establishing eligibility. If local *gBRCA* testing results are not available, central testing will be provided for those patients who otherwise appear to be eligible (see Section 6.2.1).
- 6A. Completed adequate breast surgery defined as:
  - The inked margins of breast conservation surgery or mastectomy must be histologically free of invasive breast cancer and ductal carcinoma in situ with the exception of the posterior margin if this margin is the pectoralis major fascia or the anterior margin if this is the dermis. Patients with resection margins positive for lobular carcinoma *in situ* are eligible.
  - Patients with breast conservation must have adjuvant radiotherapy. Patients having mastectomy may have adjuvant radiotherapy according to local policy and/or international guidelines.

NCI Version Date: 05-06-2021 59(177) NSABP B-55/BIG 6-13

6B. Completed adequate axilla surgery defined as:

Adjuvant Chemotherapy Patients:

- Sentinel lymph node biopsy alone if negative or if lymph node(s) only contain micrometastases (≤2.0 mm) OR
- Positive sentinel lymph node biopsy followed by axillary nodal dissection or radiotherapy as per local guidelines OR
- Axillary dissection

Neoadjuvant Chemotherapy Patients:

- Sentinel lymph node biopsy performed *before* neoadjuvant chemotherapy:
  - If negative or if lymph node(s) only contain micrometastases (≤2.0 mm), additional axillary surgery is not required
  - If positive, axillary node dissection or axillary nodal radiotherapy should follow completion of neoadjuvant chemotherapy
- Sentinel lymph node biopsy performed *after* neoadjuvant chemotherapy:
  - If negative, additional axillary surgery not mandated
  - If positive (micrometastases are regarded as positive), additional axillary surgery is required unless the patient is enrolled in a Phase III multicentre clinical trials proposing radiotherapy as alternative treatment of the axilla. The trial must be pre-approved by the OlympiA Executive Committee.
  - Axillary dissection
- 7. Completed at least 6 cycles of neoadjuvant or adjuvant chemotherapy containing anthracyclines, taxanes or the combination of both. Prior platinum as potentially curative treatment for prior cancer (e.g. ovarian) or as adjuvant or neoadjuvant treatment for breast cancer is allowed. (For neoadjuvant patients all chemotherapy should be delivered prior to surgery. No further cycles of chemotherapy post-surgery are allowed.)
- 8. Patients must have adequate organ and bone marrow function measured within 28 days prior to randomisation with no blood transfusions (packed red blood cells and/or platelet transfusions) in the past 28 days prior to testing for organ and bone marrow function as defined below:
  - Haemoglobin ≥10.0 g/dL
  - Absolute neutrophil count (ANC)  $\ge$ 1.5 x 10<sup>9</sup>/L

NCI Version Date: 05-06-2021 60(177) NSABP B-55/BIG 6-13

- Platelet count  $\ge 100 \times 10^9$ /L
- Total Bilirubin ≤ ULN (institutional upper limit of normal) except elevated total bilirubin <1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin
- AST (SGOT)/ALT (SGPT) ≤2.5 x ULN
- ALP < 2.5 x ULN

To rule out metastatic breast cancer, patients with screening ALT/AST or ALP above institutional upper limit of normal should have liver ultrasound, CT or MRI at any time point between diagnosis of current breast cancer and randomisation. Screening bone scan is required if ALP and/or corrected calcium level are above the institutional upper limit. (Note: PET/CT scan may be used as an alternative imaging technique).

- 9. Serum or plasma creatinine  $\leq 1.5 \text{ x ULN}$
- 10. ECOG performance status 0-1
- Women who are not postmenopausal or have not undergone a hysterectomy must have documented negative pregnancy test within 28 days prior to randomisation.

Postmenopausal is defined as one or more of the following:

- Age  $\geq$  60 yrs
- Age < 60 and amenorrheic for 1 year or more in the absence of chemotherapy and/or hormonal treatment
- Follicle stimulating hormone (FSH) and plasma estradiol levels in the postmenopausal range for women under 60
- Radiation-induced oophorectomy with last menses >1 year ago
- Bilateral oophorectomy
- \*\*Women of childbearing potential who are sexually active must agree, with their partners, to the use of two highly effective forms of contraception in combination. This should be started from the signing of the informed consent and continue, throughout the period of taking study treatment and for at least 1 month after the last dose of study drug, or they must totally/truly abstain from any form of sexual intercourse. Male patients must use a condom during treatment and for 3 months after last dose of study drug when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception (see <a href="Appendix E">Appendix E</a> for acceptable methods) if they are of childbearing potential.

- \*\*Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
- 13. Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary tumour, mandatory\*.
  - \*NOTE: For adjuvant patients, this refers to the surgical specimen; for neoadjuvant patients, both the pre-treatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required.
- 14. Patient should be randomised in the trial ideally within a maximum of 8 weeks of completion of their last treatment (surgery, chemotherapy or radiotherapy), but in no case longer than 12 weeks.

# 4.2 Exclusion criteria

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

- 1. \*\*Involvement in the planning and/or conduct of the study.
- 2. Patients who do not have deleterious or suspected deleterious *gBRCA1* and/or 2 mutations but only have *BRCA1* and/or *BRCA2* mutations that are considered to be non-detrimental (e.g., "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favour polymorphism" or "benign polymorphism" etc.).
- 3. \*\*Previous randomisation in the present study.
- 4. \*\*Evidence of metastatic breast cancer. Patient considered at high risk of having disseminated disease (i.e. those with locally advanced disease, clinical N2-3 or pathological N1-3 with the exception of pN1a in adjuvant patients) should have a CT/MRI scan of the Thorax/Abdomen/Pelvis or any other area as clinically indicated and a bone scan <u>or</u> a CT scan with bone windows at any point between diagnosis of the current breast cancer and randomisation to rule out metastatic breast cancer. (Note: PET/CT scan may be used as an alternative imaging technique and precludes the need for bone scan). Patients with screening ALT/AST or ALP above institutional upper limit of normal should have liver ultrasound, CT or MRI at any time point between diagnosis of current breast cancer and randomisation. Screening bone scan is required if ALP and/or corrected calcium level are above the institutional upper limit. (Note: PET/CT scan may be used as an alternative imaging technique).

NCI Version Date: 05-06-2021 62(177) NSABP B-55/BIG 6-13

- 5. \*\*Exposure to an investigational product within 30 days or five half lives (whichever is the longer) prior to randomisation.
- 6. \*\*Any previous treatment with a PARP inhibitor, including olaparib and/or known hypersensitivity to any of the excipients of study treatment.
- 7. \*\*Patients with second primary malignancy. **EXCEPTIONS** are:
  - o adequately treated non-melanoma skin cancer, curatively treated *in situ* cancer of the cervix, Ductal Carcinoma *in situ* (DCIS) of the breast, stage 1 grade 1 endometrial carcinoma
  - o other solid tumours and lymphomas (without bone marrow involvement) diagnosed ≥5 years prior to randomisation and treated with no evidence of disease recurrence and for whom no more than one line of chemotherapy was applied.
- 8. Resting ECG with QTc >470 msec detected on 2 or more time points within a 24 hour period or family history of long QT syndrome. If ECG demonstrates QTc >470 msec, patient will be eligible only if repeat ECG demonstrates QTc ≤470 msec.
- 9. Patients receiving systemic chemotherapy within 3 weeks prior to randomisation.
- 10. Patients receiving adjuvant radiotherapy within 2 weeks prior to randomisation.
- 11. Concomitant use of known strong CYP3A4 inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks. Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafmil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
- 12. Persistent toxicities (≥CTCAE grade 2) caused by previous cancer therapy, excluding alopecia and CTCAE grade 2 peripheral neuropathy.
- 13. \*\* Patients with current or past history of haematologic malignancies and any clonal non-malignant haematological disorder which predisposes the patient to develop a haematological malignancy. Exception: lymphoma (refer to Exclusion Criterion 7).
- 14. Major surgery within 2 weeks prior to randomisation: patients must have recovered from any effects of any major surgery.
- 15. Patients considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.

NCI Version Date: 05-06-2021 63(177) NSABP B-55/BIG 6-13

Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, extensive bilateral lung disease on High Resolution Computed Tomography scan or any psychiatric disorder that prohibits obtaining informed consent.

- 16. \*\*Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
- 17. Pregnant or breastfeeding women.
- 18. \*\*Patients with known active Hepatitis B or C
- 19. \*\*Patients known to be HIV positive with one or more of the following:
  - a. Baseline CD4 count of < 250 cells/mm<sup>3</sup>
  - b. History of AIDS indicator conditions
  - c. Anti-retroviral therapy with any potent CYP3A4 inhibitor (see Section 5.6.2)
- 20. \*\*Previous allogeneic bone marrow transplant.
- 21. \*\*Whole blood transfusions in the last 120 days prior to entry to the study which may interfere with *gBRCA* testing (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no. 8)

For procedures for withdrawal of incorrectly enrolled patients see <u>Section 5.3</u>.

# 5. STUDY CONDUCT

# 5.1 Restrictions during the study

#### 5.1.1 Meals and dietary restrictions

It is prohibited to consume grapefruit juice while on study therapy.

# 5.1.2 Contraception

Women of childbearing potential who are sexually active, must agree, to the use of two highly effective forms of contraception in combination (as described in <u>Appendix E</u>). This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug, or they must totally/truly abstain from any form of sexual intercourse. Male patients must use a condom during treatment and for 3 months after the last dose of study drug when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking olaparib and for 3 months following the last dose of olaparib. For details please refer to <u>Appendix E</u> Acceptable Birth Control Methods.

NCI Version Date: 05-06-2021 64(177) NSABP B-55/BIG 6-13

# 5.2 Patient enrolment and randomisation and initiation of study treatment

The following section outlines procedures for Screening Registration and for Randomisation, and for ordering Study Drug at randomisation.

- The Investigator must obtain signed informed consent from the potential patient before any study specific procedures are performed.
- Patients will be assigned a unique patient identifier (E-code) which should be used to
  identify the patient on the central Myriad sample, the eCRFs in Medidata RAVE and
  any other trial-related communications.
- 3. The Investigator must determine patient eligibility. See <u>Sections 4.1</u> and <u>4.2</u>.
- 4. If the patient meets the eligibility requirements, the authorized site staff should randomise the patient using OPEN, answering all questions which are asked by the system including questions relative to the stratification factors.
- 5. OPEN will randomly assign treatment (olaparib or placebo). The treatment allocation will be blinded for the Investigator and the patient.
- 6. Randomisation will automatically trigger study drug shipment to the site (except for countries where the initial drug shipment is sent upon activation). Details of drug ordering procedures can be found in <u>Section 5.5.5</u>.
- Once medication is received, the site personnel can then dispense the medication kit per patient's treatment assignment.

# 5.2.1 CTEP registration procedures

Food and Drug Administration (FDA) regulations and National Cancer Institute (NCI) policy require all individuals contributing to NCI-sponsored trials to register and to renew their registration annually. To register, all individuals must obtain a Cancer Therapy Evaluation Program (CTEP) Identity and Access Management (IAM) account (<a href="https://ctepcore.nci.nih.gov/iam">https://ctepcore.nci.nih.gov/iam</a>). In addition, persons with a registration type of Investigator (IVR), Non-Physician Investigator (NPIVR), or Associate Plus (AP) (i.e., clinical site staff requiring write access to OPEN, RAVE, or TRIAD or acting as a primary site contact) must complete their annual registration using CTEP's web-based Registration and Credential Repository (RCR) (<a href="https://ctepcore.nci.nih.gov/rcr">https://ctepcore.nci.nih.gov/rcr</a>). Documentation requirements per registration type are outlined in the table below.

| Documentation Required | IVR | NPIVR | AP | A |
|------------------------|-----|-------|----|---|
| FDA Form 1572 | v | > | | |

NCI Version Date: 05-06-2021 65(177) NSABP B-55/BIG 6-13

| Documentation Required | IVR | NPIVR | AP | A |
|---|---|---|---|---|
| Financial Disclosure Form | ~ | • | • | |
| NCI Biosketch (education, training, employment, license, and certification) | • | • | ¥ | |
| HSP/GCP training | ¥ | • | ¥ | |
| Agent Shipment Form (if applicable) | ¥ | T. | | |
| CV (optional) | ¥ | • | ¥ | |

An active CTEP-IAM user account and appropriate RCR registration is required to access all CTEP and CTSU (Cancer Trials Support Unit) websites and applications. In addition, IVRs and NPIVRs must list all clinical practice sites and IRBs covering their practice sites on the FDA Form 1572 in RCR to allow the following:

- Added to a site roster
- Assigned the treating, credit, consenting, or drug shipment (IVR only) tasks in OPEN
- · Act as the site-protocol PI on the IRB approval

Additional information can be found on the CTEP website at < <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a>>. For questions, please contact the RCR *Help Desk* by email as < RCRHelpDesk@nih.gov >.

# 5.2.2 CTSU registration procedures

This study is supported by the NCI Cancer Trials Support Unit (CTSU).

# 5.2.2.1 IRB approval

Each investigator or group of investigators at a clinical site must obtain IRB approval for this protocol and submit IRB approval and supporting documentation to the CTSU Regulatory Office before they can be approved to enroll patients. Assignment of site registration status in the CTSU Regulatory Support System (RSS) uses extensive data to make a determination of whether a site has fulfilled all regulatory criteria including but not limited to the following:

- An active Federal Wide Assurance (FWA) number
- An active roster affiliation with the Lead Network or a participating organization
- A valid IRB approval
- Compliance with all protocol-specific requirements.

Sites participating on the NCI CIRB initiative that are approved by the CIRB for this study are not required to submit IRB approval documentation to the CTSU Regulatory Office. For sites using the CIRB, IRB approval information is received from the CIRB and applied to the RSS in an automated process. Signatory Institutions must submit a Study Specific Worksheet for Local Context (SSW) to the CIRB via IRB Manager to indicate their intent to open the study locally. The CIRB's approval of the SSW is then communicated to the CTSU Regulatory Office. In order for the SSW approval to be processed, the Signatory Institution must inform the CTSU which CIRB-approved institutions aligned with the Signatory Institution are participating in the study.

# **5.2.2.2** Downloading site registration documents

Site registration forms may be downloaded from the NSABP B-55 protocol page located on the CTSU Members' website.

- Go to <a href="https://www.ctsu.org">https://www.ctsu.org</a> and log in to the Members' area using your CTEP-IAM username and password
- Click on the Protocols tab in the upper left of your screen
- Either enter the protocol # in the search field at the top of the protocol tree, or
- Click on the By Lead Organization folder to expand
- Click on the NRG link to expand, then select trial protocol NSABP B-55
- Click on LPO Documents, select the Site Registration documents link, and download and complete the forms provided

# 5.2.2.3 Requirements for B-55/6-13 site registration

IRB approval (For sites not participating via the NCI CIRB; local IRB documentation, an IRB-signed CTSU IRB Certification Form, Protocol of Human Subjects Assurance Identification/IRB Certification/Declaration of Exemption Form, or combination is accepted)

# **5.2.2.4** Submitting regulatory documents

Submit completed forms and documents to the CTSU Regulatory Office via the Regulatory Submission Portal, where they will be entered and tracked in the CTSU RSS.

<u>Regulatory Submission Panel</u>: <u>www.ctsu.org</u> (Members' area) → Regulatory Tab → Regulatory Submission

When applicable, original documents should be mailed to: CTSU Regulatory Office 1818 Market Street, Suite 3000 Philadelphia, PA 19103

Institutions with patients waiting that are unable to use the Portal should alert the CTSU Regulatory Office immediately at 1-866-651-2878 in order to receive further instruction and support.

#### 5.2.2.5 Checking your site's registration status

You can verify your site registration status on the Members' section of the CTSU website.

- Go to <a href="https://www.ctsu.org">https://www.ctsu.org</a> and log in to the Members' area using your CTEP-IAM username and password
- Click on the Regulatory tab
- Click on the Site Registration tab
- Enter your 5-character CTEP Institution Code and click on Go

Note: The status given only reflects compliance with IRB documentation and institutional compliance with protocol-specific requirements outlined by the Lead Network. It does not reflect compliance with protocol requirements for individuals participating on the protocol or the enrolling investigator's status with the NCI or their affiliated networks.

#### 5.2.3 Procedures for randomisation

Patient eligibility must be established before randomisation is undertaken. Randomisation can be performed for patients who met all eligibility criteria upon completion of all necessary Screening PART 2 procedures to ensure that the study drug is available at site and can be dispensed to the patient preferably during Visit 2 (Day 1).

The randomisation system will use the following stratification factors:

- Hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC)
   NOTE: In cases of multifocal, multicentric or synchronous bilateral invasive disease, stratification is based on the status of the lesion considered at highest risk (at the investigator's discretion) that was used to determine eligibility.
- Neoadjuvant versus adjuvant chemotherapy
- Platinum therapy for current breast cancer: Yes/No

Eligible patients will be randomised in a 1:1 ratio to one of the following treatments:

- Olaparib tablets p.o. 300 mg twice daily
- Matching placebo tablets p.o. twice daily

It is recommended that patients commence study treatment within 7 days of randomisation, but no later than 21 days.

If, following randomisation, it is discovered that incorrect information on the stratification factors was entered at randomisation, then the correct information should be recorded in the eCRF but the randomisation system will retain the information that was provided at the time of randomisation. The NRG Oncology SDMC must also be notified.

#### 5.2.4 Oncology Patient Enrollment Network (OPEN)

Patient enrollment will be facilitated using the Oncology Patient Enrollment Network (OPEN). OPEN is a web-based registration system available on a 24/7 basis. To access OPEN, the site

NCI Version Date: 05-06-2021 68(177) NSABP B-55/BIG 6-13

user must have an active CTEP-IAM account (check at < <a href="https://ctepcore.nci.nih.gov/iam">https://ctepcore.nci.nih.gov/iam</a> ) and a 'Registrar' role on either the LPO or participating organization roster. Registrars must hold a minimum of an AP registration type.

All site staff will use OPEN to enroll patients to this study. It is integrated with the CTSU Enterprise System for regulatory and roster data and, upon enrollment, initializes the patient in the Rave database. OPEN can be accessed at <a href="https://open.ctsu.org">https://open.ctsu.org</a> or from the OPEN tab on the CTSU Members' side of the website at <a href="https://www.ctsu.org">https://www.ctsu.org</a>. To an assign an IVR or NPIVR as the treating, crediting, consenting, drug shipment (IVR only), or investigator receiving a transfer in OPEN, the IVR or NPIVR must list on their FDA 1572 in RCR the IRB number used on the site's IRB approval.

Prior to accessing OPEN site staff should verify the following:

- All eligibility criteria have been met within the protocol stated timeframes. Site staff should use the registration forms provided on the NRG Oncology or CTSU Web site as a tool to verify eligibility.
- All patients have signed an appropriate consent form and HIPAA authorization form (if applicable).

Note: The OPEN system will provide the site with a printable confirmation of registration, including the Patient ID number for the study, and treatment information. Please print this confirmation for your records. Additionally, a transmittal form to be used when faxing the signed consent form to the NRG Oncology SDMC will be provided. If it is necessary to reprint the randomization confirmation or the transmittal form, they can be reprinted through Coordinator Online via the *View a Patient Entry Report* under Patient Entry.

Further instructional information is provided on the OPEN tab of the CTSU Member side of the CTSU Web site at <a href="https://www.ctsu.org">https://www.ctsu.org</a> or at <a href="https://open.ctsu.org">https://open.ctsu.org</a>. For any additional questions contact the CTSU Help Desk at 1-888-823-5923 or <a href="test-attention">test-attention</a> or <a href="test-attention">test-attention</a> (westat.com).

# 5.3 Procedures for handling patients incorrectly enrolled or randomised or initiated on study treatment

Patients who fail to meet the inclusion/exclusion criteria must not, under any circumstances, be enrolled or receive study medication. There can be no exceptions to this rule.

Where patients that do not meet the eligibility criteria are randomised in error or incorrectly started treatment, or where patients are subsequently found not to meet the pre-study criteria, a discussion should occur between the Protocol Officer or a Protocol Chair, if the Protocol Officer is not available (see Section 13.1), and the Investigator regarding whether to continue or discontinue the patient from treatment. Once a decision is made, Investigators need to ensure they comply with all applicable requirements for human patient protection and ethical review. The data on these patients will remain in the study database and will be included in appropriate analyses as defined by the Statistical Analysis Plan. Data values provided at the time of randomisation will not be changed. Any corrected values for stratification fields or other randomisation data fields will be recorded elsewhere in the clinical database, leaving the randomisation record to reflect the data actually provided at the time of randomisation.

NCI Version Date: 05-06-2021 69(177) NSABP B-55/BIG 6-13

Contact with the Protocol Officer or a Protocol Chair is to ensure all such decisions are appropriately documented. The NRG Oncology SDMC must also be notified. In situations where an agreement cannot be reached, the patient should have their study therapy stopped but should continue to have efficacy assessments as per the study plan, unless the patient withdraws consent.

# 5.4 Blinding and procedures for unblinding the study

# 5.4.1 Methods for ensuring blinding

Olaparib and placebo treatment will be blinded.

The active and placebo tablets will be identical and presented in the same packaging to ensure blinding of the study medication.

# 5.4.2 Methods for unblinding individual patients

The treatment code for an individual patient should not be broken except in medical emergencies and when the appropriate management of the patient requires knowledge of the actual treatment assignment. Following emergency unblinding the investigator should report the unblinding to the Protocol Officer (see Section 13.1), without revealing any treatment information.

Only life-threatening situations should be considered as emergency such as in the cases listed below:

- Study drug was taken by someone else other than the patient by mistake.
- Patient is in a life-threatening condition following intentional or unintentional consumption of study drug in higher doses than indicated.
- Patient admitted to emergency unit with what is regarded as life threatening condition irrespective of potential causal relationship with OLYMPIA study drug, and the treating team has to know the nature of all medications the patient is receiving.

Most other situations not mentioned above are regarded as non-emergency and hence the non-emergency unblinding procedure should apply.

Where a non-emergency unblinding is sought for an individual patient the process will require a discussion with the Protocol Officer (see <u>Section 13.1</u>) to understand the need for unblinding and help minimise any unnecessary unblinding, before the patient is unblinded. However, the final decision as to whether or not to unblind the patient will be made by the Investigator.

Disease progression or medical conditions that are manageable without any compromise to patient care in the absence of knowledge of the treatment received by the patient will not be considered as valid reasons for unblinding.

In both emergency and non-emergency cases, the information on the assigned treatment (i.e. Olaparib or Placebo) should be restricted only to the Principal Investigator and/or personnel involved in the clinical care of the patient as deemed appropriate by the Principal Investigator. This information should not be revealed to the monitor, sponsor or any member of the study team.

NCI Version Date: 05-06-2021 70(177) NSABP B-55/BIG 6-13

Any patient unblinded will need to be immediately discontinued from the study treatment.

The AstraZeneca patient safety team retains the right to break the code for individual SAEs that are unexpected and are suspected to be causally related to the study treatment and that potentially require expedited reporting to regulatory authorities. Treatment codes will not be broken for the planned analyses of data until all decisions on the evaluability of the data from each individual patient have been made and documented and the target number of events has been reached.

#### 5.4.3 Procedures for unblinding

When unblinding is required, local investigators must telephone the NRG Oncology SDMC (see <u>Information Resources</u>) and state that they wish to unblind a patient's study drug assignment. The same procedure applies to 24-hour emergency unblinding. A data file is maintained for the study and can be accessed by a limited number of designees within the NRG Oncology SDMC who serve the study in an administrative, nonclinical capacity. NRG Oncology SDMC personnel will require the protocol number (i.e., NSABP B-55/BIG 6-13), the patient ID number (e.g., "E999999"), the patient initials (e.g., "LFM"), and the reason for the unblinding request in order to unblind the study drug assignment. After the confirmation of the indication for unblinding is obtained, the NRG Oncology investigator will be notified immediately of the patient's treatment assignment. A computer record will be created to identify the patient as having been unblinded. The institution is responsible for providing continued follow-up (for patients whose treatment assignment has been unblinded) on the same schedule as indicated in the study protocol for patients who have not been unblinded, unless otherwise specified.

#### 5.5 Treatments

#### 5.5.1 Identity of study treatment

AstraZeneca's Pharmaceutical Development, R&D Supply Chain will supply olaparib and matching placebo to the Pharmaceutical Management Branch (PMB), Cancer Therapy Evaluation Program (CTEP), Division of Cancer Treatment and Diagnosis (DCTD), National Cancer Institute (NCI) as green film-coated tablets as shown in <u>Table 4</u> below.

 Table 4
 Identity of study treatment

| Study treatment | Dosage form and strength |
|---------------------------|---------------------------------|
| Olaparib* | Tablet -100 mg |
| Olaparib* | Tablet – 150 mg |
| Placebo to match olaparib | Tablet to match 100 mg olaparib |
| Placebo to match olaparib | Tablet to match 150 mg olaparib |

<sup>\*</sup> Descriptive information for olaparib can be found in the Investigator's Brochure

#### 5.5.2 Doses and treatment regimens

#### 5.5.2.1 Olaparib and matching placebo (study treatment)

The planned dose of 300 mg b.i.d. (twice daily) will be made up of two (2) x 150 mg tablets b.i.d. (twice daily) with 100 mg tablets used to manage dose reductions as explained in <u>Table 5</u>.

Table 5 Study treatment doses and treatment regimens

| Total | <u>Dose</u> | Mor | ning | Eve | ning |
|---|---|---|---|---|---|
| <u>daily dose</u> | twice daily<br>(b.i.d.) | Number of tablets | <u>Tablet</u><br>strength | Number of tablets | <u>Tablet</u><br>strength |
| 600 mg | 300 mg | 2 tablets | 150 mg | 2 tablets | 150 mg |
| Initial dose (3 | 00 mg twice dail | y) can be reduce | d as follows for A | AEs (no re-escala | tion allowed): |
| <b>7</b> 00 | 2.50 | 1 tablet | 150 mg | 1 tablet | 150 mg |
| 500 mg | 250 mg | 1 tablet | 100 mg | 1 tablet | 100 mg |
| 400 mg | 200 mg | 2 tablets | 100 mg | 2 tablets | 100 mg |
| Tempo | rary dose levels o | lue to CYP3A in | hibitor exposure | (re-escalation al | lowed): |
| 300 mg | 150 mg | 1 tablet | 150 mg | 1 tablet | 150 mg |
| 200 mg | 100 mg | 1 tablet | 100 mg | 1 tablet | 100 mg |

As soon as possible following randomisation, patients will be administered olaparib or matching placebo orally twice daily (b.i.d.) at 300 mg for 52 weeks. Two (2) x 150 mg olaparib or matching placebo tablets should be taken at the same time each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water. The olaparib/placebo tablets should be swallowed whole and not chewed, crushed, dissolved or divided. Olaparib/placebo tablets can be taken with a light meal/snack (e.g., two pieces of toast or two biscuits).

If vomiting occurs shortly after the study treatment tablets are swallowed, the dose should only be replaced if all of the intact tablets can be seen and counted. Should any patient enrolled on the study miss a scheduled dose for whatever reason (e.g., as a result of forgetting to take the tablets or vomiting), the patient will be allowed to take the scheduled dose up to a maximum of 2 hours after that scheduled dose time. If greater than 2 hours after the scheduled dose time, the missed dose is not to be taken and the patient should take their next allotted dose at the next scheduled time. Patients should not take two doses (4 tablets) at the same time.

Within this study, patients will not be provided olaparib post discontinuation of study treatment. Patients and investigators will not be routinely unblinded to study treatment prior to the final overall survival (OS) analysis.

#### 5.5.3 Olaparib/Placebo

#### • Chemical name

4-(3-{[4-(Cyclopropylcarbonyl)piperazin- 1 - yl]carbonyl}-4-fluorobenzyl)phthalazin-1(2H)-one

#### • Trade name

Olaparib

#### • Classification

Poly (ADP ribose) polymerase 1 inhibitor (PARPi)

# • CAS registry number

763113-22-0

# • Molecular formula

C24H23FN4O3

# • Molecular weight

434.46

## • Approximate solubility

Olaparib is a crystalline solid. Olaparib is non-chiral. Olaparib shows pH-independent solubility across the physiological range of approximately 0.1 mg/ml.

### Mode of action

Olaparib (AZD2281, KU-0059436) is a potent inhibitor of poly (ADP-ribose) polymerase enzyme (PARP) that is being developed as a monotherapy as well as well as for combination with chemotherapy, ionizing radiation, and other anti-cancer agents. Poly (ADP-ribose) polymerase inhibition is a novel approach to targeting tumors that have homologous recombination DNA repair (HRR) pathway deficiencies (HRD). In HRD tumors, single agent treatment with olaparib can lead to tumor regression by a process known as synthetic lethality – a result of the accumulation of un-repaired DNA double-strand breaks (DSB) and an unsupportable increase in genomic instability. Olaparib may also enhance the DNA damaging effects of ionizing radiation and chemotherapy.

# • Description

The 100 mg and 150 mg strengths of olaparib tablets are composed of the same constituents. The tablet cores comprise: olaparib, copovidone, colloidal silicon dioxide, mannitol, and sodium stearyl fumarate. The composition of the tablet film-coating is: hydroxypropyl methylcellulose (hypromellose), macrogol 400 (polyethylene glycol 400), titanium dioxide, iron oxide yellow, and iron oxide black.

Placebo tablets are identical in appearance to olaparib film-coated tablets. These tablets contain: mannitol, microcrystalline cellulose, sodium starch glycolate, and magnesium stearate. The composition of the film coat is identical to that of the olaparib film-coated tablet.

# How supplied

For this study, olaparib and matching placebo will be supplied by AstraZeneca and will be distributed by the Pharmaceutical Management Branch (PMB), Cancer Therapy Evaluation Program (CTEP), Division of Treatment and Diagnosis (DCTD), National Cancer Institute (NCI).

NCI Version Date: 05-06-2021 73(177) NSABP B-55/BIG 6-13

Olaparib is presented as a green, film-coated tablet containing 100 mg or 150 mg of drug substance. The placebo tablets do not contain the active drug substance. Both the olaparib and matching placebo tablets are supplied in high-density polyethylene (HDPE) bottles. Each bottle will contain 32-150 mg or 100 mg tablets (olaparib 150 mg or 100 mg) or 0 mg tablets (placebo for olaparib 150 mg or 100 mg) and a desiccant. Bottles are secured with a child-resistant closure; induction-sealed membranes provide tamper evidence.

Olaparib and matching placebo tablets will be distributed in kits. Each kit will consist of a small box containing 2 bottles of olaparib or placebo tablets. Both bottles and kit box will contain patient-specific labels (Section 5.5.11). Each kit will contain a 16 day supply of olaparib or placebo.

- Each 300 mg kit will contain 2 bottles of olaparib or placebo 150 mg tablets
- Each 250 mg kit will contain 1 bottle of olaparib or placebo 100 mg tablets and
   1 bottle of olaparib or placebo 150 mg tablets
- Each 200 mg kit will contain 2 bottles of olaparib or placebo 100 mg tablets

# • Storage

All study drugs should be kept in a secure place under appropriate storage conditions. The investigational product label on the bottle specifies the appropriate storage.

#### • Route of administration

Oral

# Method of administration

The olaparib/placebo tablets should be swallowed whole and not chewed, crushed, dissolved, or divided. Olaparib/placebo tablets can be taken with a light meal/snack.

#### • Stability

Bottle contents are to be discarded 90 days after the seal is broken. Investigators will be notified when lots have expired.

# • Patient care implications

Pre-clinical data indicate that olaparib can have adverse effects on embryofoetal survival and development. It is not known whether olaparib is excreted in human milk. Therefore, olaparib must not be used during pregnancy or breast-feeding, and patients of childbearing potential must use contraception.

Refer to Appendix E: Acceptable Birth Control Methods for more information.

# 5.5.3.1 Drug information

Please refer to <u>Section 5.5.2</u> for study treatment and the current FDA-approved Investigator's Brochure and the site-specific pharmacy for toxicity information and instructions for drug preparation, handling, and storage.

NCI Version Date: 05-06-2021 74(177) NSABP B-55/BIG 6-13

# 5.5.4 Obtaining an Investigator's Brochure

Please refer to the current Investigator's Brochure for detailed information regarding olaparib. The olaparib IB can be downloaded from the Members' Area of the NSABP Web site or requested from the CTSU using the CTSU Request for Clinical Brochure Form posted on the CTSU Web site.

# 5.5.5 Procurement of olaparib (IND #122443, NSC #747856)/placebo

Olaparib (NSC #747856) and matching placebo will be supplied free of charge by AstraZeneca, and will be distributed by the Pharmaceutical Management Branch (PMB), Division of Cancer Therapy Treatment and Diagnosis (DCTD), National Cancer Institute (NCI). PMB policy requires that olaparib/placebo be shipped directly to the institution where the patient is to be treated.

Study supplies are packaged in "kits." Each kit contains 2 bottles of olaparib or matching placebo tablets. The label instructions on each bottle read "Take 1 tablet by mouth twice a day." This consistency of dosing instructions among dose levels is intended to avoid dosing errors for patients receiving 250 mg.

Note: Kits are to be dispensed intact. Do not separate the bottles. Instruct patients to take 1 tablet from each bottle in the kit twice a day.

No blinded starter olaparib/placebo will be available for this study. Blinded, patient-specific olaparib/placebo will be sent to the registering investigator at the time of randomisation and should arrive within approximately 5 business days. Once a patient has been randomised, the NRG Oncology SDMC will electronically transmit a clinical drug request for that patient to the PMB. The request will be processed by the PMB the next business day and shipped the following business day. Shipments will be sent by FedEx Ground (up to 5 business days for delivery but can be expedited by the provision of an express courier account name and number to the NRG Oncology SDMC at the time the patient is randomised. Please note that additional processing time is required for QA/QC checks on patient-specific/blinded orders and next day delivery is not available.

The initial shipment will contain 8 kits (16 bottles) of olaparib or placebo, enough olaparib or placebo to complete 16 weeks of therapy (2 tablets twice a day for 28 days per cycle).

Subsequent orders for blinded, patient-specific supplies must be requested by the Principal Investigator (or his/her authorized designee[s]) for NSABP B-55/BIG 6-13 at each participating institution using the PMB On-line Agent Order Processing (OAOP) program. The assigned patient ID number (e.g., E999999) and the patient initials (e.g., "LFM") should be entered in the "Patient or Special Code" field. A separate order is required for each patient ID number (e.g., E999999) being ordered. All drug orders should be shipped directly to the physician responsible for treating the patient. Requests can be placed 12 weeks after the last shipment is received. It is recommended that 6 kits (12 bottles) be requested at each order. The recommended ordering schedule is Weeks 11, 23, and 35.

Pharmaceutical Management Branch (PMB) policy requires that agent be shipped directly to the institution where the patient is to be treated. PMB does not permit the transfer of agents between institutions (unless prior approval from PMB is obtained). The CTEP-assigned protocol number must be used for ordering all CTEP-supplied investigational agents. The responsible investigator

NCI Version Date: 05-06-2021 75(177) NSABP B-55/BIG 6-13
at each participating institution must be registered with CTEP, DCTD through an annual submission of FDA Form 1572 (Statement of Investigator), Curriculum Vitae, Supplemental Investigator Data Form (IDF), and Financial Disclosure Form (FDF). If there are several participating investigators at one institution, CTEP-supplied investigational agents for the study should be ordered under the name of one lead investigator at that institution.

Active CTEP-registered investigators and investigator-designated shipping designees and ordering designees must submit agent requests through the PMB Online Agent Order Processing (OAOP) application. Access to OAOP requires the establishment of a CTEP Identity and Access Management (IAM) account and the maintenance of an "active" account status and a "current" password. For questions about drug orders, transfers, returns, or accountability, call or email PMB at any time. Refer to the PMB's website for specific policies and guidelines related to agent management.

# 5.5.6 Special ordering procedures for patients requiring a dose reduction

If the patient is **dose reduced** from 300 mg b.i.d. to 250 mg b.i.d. (or 250 mg b.i.d. to 200 mg b.i.d.), an agent request must be submitted by the site through the OAOP application.

- For each 250 mg kit, request 1 bottle of 100 mg tablets and 1 bottle of 150 mg tablets.
- For each 200 mg kit, request 2 bottles of 100 mg tablets.

The number of kits included in the initial shipment will depend on the patient's place on the treatment calendar.

# 5.5.7 Agent inventory records

The investigator, or a responsible party designated by the investigator, must maintain a careful record of the receipt, dispensing and final disposition of all agents received from the PMB using the appropriate NCI Investigational Agent (Drug) Accountability Record (DARF) available on the CTEP forms page. Store and maintain separate NCI Investigational Agent Accountability Records for each agent, strength, formulation and ordering investigator on this protocol.

#### 5.5.8 Useful Links and Contacts

- CTEP Forms, Templates, Documents: <a href="http://ctep.cancer.gov/forms/">http://ctep.cancer.gov/forms/</a>
- NCI CTEP Investigator Registration: <a href="mailto:PMBRegPend@ctep.nci.nih.gov">PMBRegPend@ctep.nci.nih.gov</a>
- PMB policies and guidelines: http://ctep.cancer.gov/branches/pmb/agent\_management.htm
- PMB Online Agent Order Processing (OAOP) application: https://ctepcore.nci.nih.gov/OAOP
- CTEP Identity and Access Management (IAM) account: https://eapps-ctep.nci.nih.gov/iam/
- CTEP Associate Registration and IAM account help: ctepreghelp@ctep.nci.nih.gov
- PMB email: PMBAfterHours@mail.nih.gov
- PMB phone and hours of service: (240) 276-6575 Monday through Friday between 8:30 am and 4:30 pm (ET)

# 5.5.9 Transfer of olaparib/placebo

Kits/bottles may *not* be transferred from one patient to another patient or from one protocol to another protocol. PMB does not permit the transfer of agents between institutions (unless prior

approval from PMB is obtained). Olaparib/placebo may not be used outside the scope of this protocol, nor can olaparib/placebo be transferred or licensed to any party not participating in this clinical study. To obtain an approval for transfer, investigators should complete and submit to the PMB (fax number 240-276-7893) a Transfer Investigational Agent Form available on the NCI home page (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>) or call the PMB at 240-276-6575. The participating institution should also inform the NRG Oncology SDMC of the transfer.

#### 5.5.10 Return of olaparib/placebo

At the completion of accrual and treatment, all unused (unopened) bottles of olaparib/placebo must be returned to the PMB. When it is necessary to return study drug (e.g., unused bottles remaining when the protocol is closed to accrual and treatment at a participating clinical site or unopened expired bottles), investigators should return the olaparib/placebo to the PMB using the NCI Return Agent Form available on the NCI home page (http://ctep.cancer.gov) or call the PMB at 240-276-6575.

Tablets remaining from dispensed bottles should be documented on the patient-specific NCI Investigational Agent Accountability Record Form for Oral Agents. On the correct dispensing row, document the date returned and the quantity, then destroy on site in accordance with institutional policy.

# 5.5.11 Labelling

For **BLINDED** (olaparib or placebo) **THERAPY**, each bottle will be labeled with:

- the protocol number (i.e., "NSABP-B-55")
- the bottle number (i.e., "Bottle 1 of 2, 2 of 2")
- the number of tablets (i.e., "32 tablets")
- the patient ID number (e.g., "E999999", where "E999999" represents a unique patient identifier assigned by NRG Oncology at registration)
- the patient initials (i.e., last initial, first initial, middle initial [e.g., "L, FM"])
- the agent identification (i.e., "Olaparib 150 mg or Placebo")
- a blank line for the pharmacist to enter the patient's name
- administration instructions (i.e., "Take <u>1</u> tablet by mouth twice a day. Discard contents after 90 days")
- storage instructions (i.e., "Store below 30°C (86°F).")
- emergency contact instructions
- a Julian date

The Julian date indicates the day the bottle was labeled and shipped and is composed of the last two digits of the calendar year (e.g., 2013 = 13, 2014 = 14) and a day count (e.g., January 1 = 001, December 31 = 365). For example, a bottle labeled and shipped on January 1, 2013, would have a Julian date of '13001' and a bottle labeled and shipped on December 31, 2014, would have a Julian date of '14365'. The Julian date will be used by PMB for recalls. When a lot expires,

NCI Version Date: 05-06-2021 77(177) NSABP B-55/BIG 6-13

PMB will determine the last date the expired lot was shipped and will recall all bottles (i.e., both Olaparib and Placebo) shipped on or before that date thus eliminating any chance of breaking the blind. The combination Julian Date – Order Number, located in the in the upper right hand corner of the bottle label, should be recorded in the lot number field on the Oral DARF.

# Each BLINDED (olaparib or placebo) KIT BOX will be labeled with:

- the protocol number (i.e., "NSABP-B-55")
- the patient ID number (e.g., "E999999", where "E999999" represents a unique patient identifier assigned by NRG Oncology at registration)
- the patient initials (i.e., last initial, first initial, middle initial [e.g., "L, FM"])
- the agent identification (i.e., "Olaparib 300 mg or Placebo Kit")
- a blank line for the pharmacist to enter the patient's name
- administration instructions (i.e., "Take 1 tablet from each bottle twice a day.")
- storage instructions (i.e., "Store below 30°C (86°F).")
- emergency contact instructions
- a Julian date

# 5.5.12 Management of toxicity of study treatment

#### **General instructions**

- The CTCAE v4.0 must be used to grade the severity of AEs.
- All dose modifications should be based on the AE requiring the greatest modification.
- Therapy should be held until the AE returns to ≤ grade 1 unless specified otherwise in the dose modification instructions.
- If study drug must be held for more than 4 weeks due to an AE or for any other reasons, permanently discontinue olaparib/placebo.
- Once a dose has been reduced, dose escalation is not permitted.
- If olaparib/placebo must be permanently discontinued, patient follow-up continues to be required as described on Table 2 and Table 3.
- If any investigational treatment is administered, olaparib/placebo must be discontinued.

# 5.5.12.1 Study therapy following breast cancer recurrence or second primary cancer

Olaparib/placebo must be discontinued following diagnosis of breast cancer recurrence or diagnosis of a second primary malignancy (i.e., excluding new in situ carcinomas of any site and squamous or basal cell skin cancers). Further therapy is at the investigator's discretion.

# 5.5.12.2 Olaparib/placebo dose levels

All olaparib/placebo dose reductions are based on the dose levels listed in Table 6.

NCI Version Date: 05-06-2021 78(177) NSABP B-55/BIG 6-13

Any toxicity observed during the course of the study should be managed by guidelines as outlined in <u>Table 7 Table 8 and Table 9</u>. Once a dose has been reduced, dose re-escalation to a higher dose is not permitted.

Table 6 Olaparib/placebo dose levels

| | Dose Level (mg) twice daily | | | | |
|---|---|---|---|---|---|
| | Starting Dose | Dose levels for AEs (no re-escalation) | | Temporary dose levels due to CYP3A inhibitor exposure | |
| Olaparib/placebo | 300 | 250 | 200 | 150 | 100 |

Table 7 Mandatory treatment for hematologic toxicity and treatment guidance for other olaparib/placebo toxicities

# **Important table instructions:**

| • Dose modifications must be based on the AE requiring the greatest modification. | | | |
|---|---|---|---|
| | Adverse Event | CTCAE<br>(v 4.0)<br>Grade | Action to be Taken |
| | Anaemia | 2<br>(8.0-9.5<br>g/dL) | Hold study therapy until > 9.5 g/dL: If recovery without packed red blood cells transfusion takes: 1-2 weeks – maintain dose; 3-4 weeks – ↓ one dose level If packed red blood cells transfusion given: reduce one dose level |
| Hematologic<br>Toxicity | | 3, 4 | Hold study therapy until > 9.5 g/dL:<br>$1^{st}$ appearance $-\downarrow 1$ dose level<br>$2^{nd}$ appearance $-\downarrow 2$ dose levels or discontinuation |
| Mandatory | Neutrophil count<br>decreased<br>(incl. febrile<br>neutropenia) | 3 | Hold study therapy until ≥ 1200/mm <sup>3</sup> ↓ one dose level |
| | | 4 | Hold study therapy until ≥ 1200/mm <sup>3</sup> ↓ two dose levels |
| | Platelet count decreased | 2 | Hold study therapy until ≥ 75,000//mm <sup>3</sup> $\downarrow$ one dose level |
| | | 3,4 | Hold study therapy until ≥ 75,000//mm <sup>3</sup> ↓ two dose levels |
| Other toxicity deemed to be attributable to study | Diarrhea (if attributable to olaparib/placebo) | 2 | Maintain dose or ↓ one dose level |
| | | 3 | ↓ one dose level |
| | | 4 | Discontinuation |
| treatment | Mucositis – oral | 2 | Maintain dose or ↓ one dose level |
| Guidance | | 3 | ↓ one dose level |
| | | 4 | Discontinuation |

Table 7 Mandatory treatment for hematologic toxicity and treatment guidance for other olaparib/placebo toxicities

# **Important table instructions:**

• Dose modifications must be based on the AE requiring the greatest modification.

| 1 8 8 | | | |
|---|---|---|---|
| | Adverse Event | CTCAE<br>(v 4.0)<br>Grade | Action to be Taken |
| | Nausea (despite antiemetics) | 2 | Maintain dose or ↓ one dose level |
| | | 3 | ↓ one dose level |
| | Vomiting (despite antiemetics) | 2 | Maintain dose or ↓ one dose level |
| | | 3 | ↓ one dose level |
| | | 4 | ↓ one dose level or discontinuation |
| Other toxicity deemed to be attributable to study treatment Guidance | Infection | 3 | Hold study therapy: When resolved: Maintain dose or ↓ one dose level Repeat appearance – ↓ one dose level |
| | | 4 | Hold study therapy: When resolved: ↓ two dose levels or discontinuation |
| | Dyspnea | 1, 2, 3 | Hold study therapy; rule out pneumonitis Follow instructions in footnote <b>a</b> |
| | | 4 | Discontinuation |
| | Pneumonitis | 2 | Follow instructions in footnote a |
| | | 3, 4 | Discontinuation |
| | Other clinically significant AEs deemed related to | 2 | Maintain dose or ↓ one dose level |
| | | 3 | ↓ one dose level |
| | study treatmentb | 4 | ↓ two dose levels or discontinuation |

a Hold olaparib/placebo and determine etiology. Unless prohibited based on instructions for other clinical diagnoses (i.e. other AEs), resume olaparib/placebo when grade 0 (if the AE requiring olaparib to be held was dyspnea) or when ≤ grade 1 (if the AE requiring olaparib/placebo to be held was ≥ grade 2).

Table 8 Dose reduction for study treatment to manage moderate renal impairment

| Initial dose | Moderate renal impairment (calculated creatinine clearance<br>by Cockcroft -Gault equation or based on a 24 hour urine<br>test between 31 and 50 ml/min): Dose reduction |
|---|---|
| 300 mg twice daily | 200 mg twice daily |

b Determination of "clinically significant" AEs is at the investigator's discretion.

Table 9 Dose reduction for study treatment with concurrent use of a strong or moderate CYP3A inhibitor

| Initial dose | Strong CYP3A inhibitor | Moderate CYP3A inhibitor |
|--------------------|------------------------|--------------------------|
| 300 mg twice daily | 100 mg twice daily | 150 mg twice daily |

For guidance on dose reductions for management of renal impairment refer to Section 5.5.12.3,

For guidance on dose reductions when concomitant strong or moderate CYP3A inhibitors cannot be avoided see section 5.6.2.

# 5.5.12.3 Renal impairment

If subsequent to study entry and while still on study therapy, a patient's estimated creatinine clearance falls below the threshold for study inclusion (>51 ml/min), retesting should be performed promptly.

A dose reduction is recommended for patients who develop moderate renal impairment (calculated creatinine clearance by Cockcroft-Gault equation or based on a 24 hour urine test of between 31 and 50 ml/min) for any reason during the course of the study: the dose of study treatment should be reduced to 200 mg b.i.d.

Because the creatinine clearance determination is only an estimate of renal function, in instances where the creatinine clearance falls between 31 and 50 mL/min, the investigator should use his or her discretion in determining whether a dose change or discontinuation of therapy is warranted.

Olaparib has not been studied in patients with severe renal impairment (creatinine clearance <30 ml/min) or end-stage renal disease; if patients develop severe impairment or end stage disease is it recommended that study treatment be discontinued.

# 5.5.12.4 Management of haematological toxicity

If blood transfusion support is required to maintain haemoglobin levels above 9.5 g/dL at Dose Level -2 with no alternative explanation for the recurring anaemia, study treatment should be permanently discontinued and the patient referred for haematological evaluation.

If a patient develops febrile neutropenia, study treatment should be stopped and appropriate management including G-CSF may be given according to local hospital guidelines. If grade 3 or 4 anaemia, neutropenia or thrombocytopenia occurs, weekly differential blood counts including reticulocytes and peripheral blood smear should be performed until Hgb is > 9.5 g/dL, ANC is > 1200/mm³ and platelets are > 75,000/mm³. If persistent haematological toxicities lead to discontinuation of study therapy, the patient should be referred to a haematologist for further investigations. Differential blood counts including reticulocytes and peripheral blood smear should be performed at least every 2 weeks until resolution or stabilization.

NCI Version Date: 05-06-2021 82(177) NSABP B-55/BIG 6-13

Bone marrow analysis and/or blood cytogenetic analysis should be considered at this stage according to standard haematological practice. Clinical notes and results from further testing should be submitted.

Development of a confirmed myelodysplastic syndrome or other clonal blood disorder should be reported as an SAE.

Administration of blood cell products and platelet transfusions must be recorded in eCRF.

# 5.5.12.5 Management of new or worsening pulmonary symptoms

If new or worsening pulmonary symptoms (e.g., dyspnoea) or radiological abnormality occurs, study treatment should be held and a diagnostic workup (including a high resolution CT scan) should be performed, to exclude pneumonitis. Following investigation, if no evidence of abnormality is observed on CT imaging and symptoms resolve, then study treatment can be restarted, if deemed appropriate by the investigator. If significant pulmonary abnormalities are identified, these need to be discussed with the Protocol Officer (see Section 13.1).

# 5.5.12.6 Management of nausea and vomiting

No routine prophylactic anti-emetic treatment is required at the start of study treatment; however, patients should receive appropriate anti-emetic treatment at the first onset of nausea or vomiting and as required thereafter, in accordance with local treatment practice guidelines. As per international guidance on antiemetic use in cancer patients (ESMO, NCCN), generally a single agent antiemetic should be considered.

# 5.5.12.7 Interruptions for intercurrent non-toxicity related events

Study treatment dose interruption for conditions other than toxicity resolution should be kept as short as possible. If a patient cannot restart study treatment within 4 weeks for resolution of intercurrent conditions not related to disease recurrence or toxicity, the case should be discussed with the Protocol Officer (see Section 13.1). All dose reductions and interruptions (including any missed doses), and the reasons for the reductions/interruptions are to be recorded according to the eCRF guidelines. Study treatment should be stopped at least 3 days prior to planned surgery. After surgery study treatment can be restarted when the wound has healed. No stoppage of study treatment is required for any needle biopsy procedure. Study treatment should be discontinued for a minimum of 3 days before a patient undergoes radiation treatment. Study treatment should be restarted within 4 weeks as long as any bone marrow toxicity has recovered. Because the AEs related to olaparib may include asthenia, fatigue and dizziness, patients should be advised to use caution while driving or using machinery if these symptoms occur.

# 5.6 Concomitant and subsequent treatment(s)

Any concomitant medications (exceptions described in <u>Table 10</u>) which are considered necessary for the patient's welfare, and which will not interfere with the study medication (in the opinion of the treating physician), may be given at the discretion of the investigator, providing the medications, the doses, dates and reasons for administration are recorded on the appropriate eCRF page in Medidata Rave.

NCI Version Date: 05-06-2021 83(177) NSABP B-55/BIG 6-13

Bisphosphonates or denosumab are allowed during study treatment phase and follow-up.

In addition, any relevant unplanned diagnostic, therapeutic or surgical procedure performed during the study period must be recorded. This includes any blood transfusions.

The reasons for the use, doses and dates of treatment should be recorded in the patient's medical records and appropriate sections of the eCRF.

All medications (prescriptions or over the counter medications) continued at the start of study or started during the study or until 30 days from the end of the last protocol treatment and different from the study medication must be documented.

Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse.

The receipt of other anti-neoplastic medications (with the exception of hormonal therapies as addressed in <u>Section 5.6.1</u>) and other investigational medication is prohibited during study treatment and follow-up.

Subsequent anti-cancer treatment is expected to be initiated following breast cancer recurrence; if subsequent anti-cancer treatment needs to be initiated during the 1-year treatment phase, study treatment must be stopped. Information on first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time must be recorded in the clinical database.

# 5.6.1 Administration of endocrine therapy

Patients should receive adjuvant endocrine therapy per local policy and/or international guidelines. Information on endocrine therapies should be collected and recorded in the eCRF until IDFS endpoint is met due to breast cancer related distant relapse.

#### 5.6.2 Restricted concomitant medications

The use of any natural/herbal products or other traditional remedies should be discouraged but use of these products, as well as any medication or vaccine including over-the-counter or prescription medicines, vitamins, and/or herbal supplements that the patient is receiving at the time of enrolment or receives during the study must be recorded along with:

- Reason for use
- Dates of administration including start and end dates
- Dosage information including dose and frequency

Table 10 Restricted concomitant medications

# Medication/class of drug: Usage (including limits for duration permitted and special situations in which it's allowed):

# Strong CYP3A inhibitors:

itraconazole, telithromycin, clarithromycin, boosted protease inhibitors, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir

#### Moderate CYP3A inhibitors:

ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil

# Strong CYP3A inducers:

phenobarbital, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine, enzalutamide and St John's Wort

#### Moderate CYP3A inducers:

bosentan, efavirenz and modafinil

Strong or moderate CYP3A inhibitors should not be taken with study treatment. If there is no suitable alternative concomitant medication then the dose of study treatment should be reduced for the period of concomitant administration. The dose reduction of study treatment should be recorded in the CRF with the reason documented as concomitant CYP3A inhibitor use.

- Strong CYP3A inhibitors reduce the dose of study treatment to 100 mg b.i.d for the duration of concomitant therapy with the strong inhibitor and for 5 halflives afterwards.
- Moderate CYP3A inhibitors reduce the dose of study treatment to 150 mg b.i.d for the duration of concomitant therapy with the moderate inhibitor and for 3 half-lives afterwards.
- After the washout of the inhibitor is complete, the study treatment dose can be re-escalated.

Strong or moderate CYP3A inducers should not be taken with study treatment.

If the use of any strong or moderate CYP3A inducers are considered necessary for the patient's safety and welfare this could diminish the clinical efficacy of olaparib.

If a patient requires use of a strong or moderate CYP3A inducer then they must be monitored carefully for any change in efficacy of study treatment.

 Table 10
 Restricted concomitant medications

| Medication/class of drug: | Usage (including limits for duration permitted and special situations in which it's allowed): |
|---|---|
| CYP3A4 substrates: hormonal | Effect of olaparib on other drugs |
| contraceptive, simvastatin, cisapride, cyclosporine, ergot alkaloids, fentanyl, pimozide, sirolimus, tacrolimus and quetiapine | Based on limited in vitro data, olaparib may increase the exposure to substrates of CYP3A4, OATPIB1, OCT1, OCT2, OAT3, MATE1 and MATE2K. |
| • CYP2B6 substrates: bupropion, efavirenz | Based on limited in vitro data, olaparib may |
| • OATP 1 B1 substrates: bosentan, | reduce the exposure to substrates of 2B6. |
| glibenclamide, repaglinide, statins and valsartan | Caution should be observed if substrates of these isoenzymes or transporter proteins are |
| • OCT1, MATE1 and MATE2K substrates: metformin | co-administered. |
| OCT2 substrates: serum creatinine | |
| • OAT3 substrates: furosemide, methotrexate | |
| Anticoagulant therapy | Patients who are taking warfarin may participate in this trial; however, it is recommended that international normalised ratio (INR) be monitored carefully at least once per week for the first month, then monthly if the INR is stable. Subcutaneous heparin and low molecular weight heparin are permitted. |
| Administration of other anti-cancer agents | Patients must not receive any other concurrent anti-cancer therapy, including investigational agents, while on study treatment. Patients may continue the use of bisphosphonates or denosumab. |

# 5.6.3 Anti-emetics/Anti-diarrheals

Should a patient develop nausea, vomiting and/or diarrhea, then these symptoms should be reported as AEs (see Section 6.4.9) and appropriate treatment given.

# 5.6.4 Live virus and bacterial vaccines

Live virus and bacterial vaccines should not be administered whilst the patient is receiving study treatment and during the 30-day follow-up period. An increased risk of infection by the

administration of live virus and bacterial vaccines has been observed with conventional chemotherapy drugs and the effects with olaparib are unknown.

# 5.7 Treatment compliance

The administration of all study drugs during the 1-year treatment phase of the study should be recorded in the appropriate sections of the eCRF.

Patients should be given clear instructions on how and when to take their study treatment. Patients will self-administer study treatment. Study site staff should do a tablet count at regular intervals during treatment. Compliance will be assessed by the tablet count and the information should be recorded in the appropriate section of the eCRF. The number of tablets returned is to be noted in the return column of the Oral Drug Accountability Record (DARF) then destroyed per the institution's standard operating procedures. All patients must return their bottle(s) of study treatment at the appropriate scheduled visit, when a new bottle will be dispensed. Patients should be instructed to notify study site personnel of missed doses. Site staff will then complete the relevant eCRF pages to document the drug actually given.

Patients should return all containers and tablets at the next scheduled visit or at the End of Treatment visit.

# 5.7.1 Accountability

The study drug provided for this study will be used only as directed in the study protocol.

The study personnel will account for all study drugs dispensed to and returned from the patient.

The investigator, or a responsible party designated by the investigator, must maintain a careful record of the receipt, disposition, and return of all olaparib/placebo received from the PMB according to good clinical practices and NCI guidelines using the NCI Investigational Agent Accountability Record for Oral Agents available on the NCI home page (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>) or by calling the PMB at 240-276-6575. Refer to the NCI Investigator's Handbook for procedures for Drug Accountability and Storage

http://ctep.cancer.gov/investigatorResources/docs/InvestigatorHandbook.pdf). Certificates of delivery, destruction and return should be signed and retained. Any discrepancies must be accounted for on the appropriate forms.

A separate Oral NCI Investigational Agent Accountability Record must be maintained for patient ID number (e.g., E999999) and tablet strength (e.g., 100 mg, 150 mg) on this protocol. The combination Julian Date – Order Number, located in the in the upper right hand corner of the bottle label, should be recorded in the lot number field on the Oral DARF.

# 5.8 Discontinuation of study treatment

Patients may be discontinued from the study treatment in the following situations:

- Patient decision. The patient is free at any time to discontinue study treatment, without prejudice to further clinical care
- Adverse Event

- Completion of 12 months treatment period
- Confirmed pregnancy during treatment
- Severe non-compliance with study protocol
- Loco-regional breast cancer recurrence (ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence)
- Distant breast cancer recurrence
- Contralateral invasive breast cancer or second primary non-breast invasive cancer
- Death
- Bone marrow findings consistent with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML)

# 5.8.1 Procedures for discontinuation of a patient from study treatment

A patient that decides to discontinue study treatment should always be asked about the reason(s) and the presence of any adverse events. If possible, he/she will be seen and assessed by an investigator(s). Adverse events will be followed up (See Sections 6.4.9 and 6.4.10); questionnaires and all study drugs should be returned by the patient.

If a patient is withdrawn from study, see <u>Section</u> <u>5.9</u>.

If patients discontinue study treatment early, the NRG Oncology SDMC must be informed immediately.

Any patient discontinuing study treatment prior to completing 52 weeks should attend the treatment discontinuation visit, if possible. Thereafter the patient should be seen at 30 days post discontinuation for the evaluations outlined in the study schedule.

After premature discontinuation of study treatment, the principal investigator/sub-investigator will continue to provide appropriate clinical care and, as far as possible, follow the study visit schedule. Only the visits where efficacy assessments are scheduled should be performed i.e., week 12, 24, 38, and 52 (as applicable) in Year 1 and all visits in Year 2 onwards. Only the following assessments should be done: recurrent/new cancers assessment, mammogram and/or breast MRI, and Quality of Life questionnaires.

Collection of vital signs, AEs, haematology/clinical chemistry results and concomitant medications is no longer required. Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse. The date of discontinuation, the reasons, and details of these specific cancer therapies (first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time) should also be recorded on the eCRF.

Samples should be collected at disease recurrence per protocol: blood biomarker samples (mandatory) and tumour sample (optional). If a recurrent/new cancer assessment is scheduled

NCI Version Date: 05-06-2021 88(177) NSABP B-55/BIG 6-13

within 4 weeks of the study treatment discontinuation visit, it can be performed at 30-day followup visit.

Patients who meet the IDFS endpoint while on study therapy should attend the treatment discontinuation visit and follow-up visit 30 days after the last dose of study treatment. See Section 3 for guidelines on subsequent study visits, which are dependent on which IDFS endpoint has been met.

After discontinuation of study treatment at any points in the study, all ongoing AEs or SAEs must be followed until resolution unless, in the investigator's opinion the condition is unlikely to resolve due to the patients underlying disease, or the patient is lost to follow-up (see Sections 6.4.9 and 6.4.10). All new AEs and SAEs occurring during the 30 calendar days after the last dose of study medication must be reported (if SAEs, they must be reported as described in Section 6.4.10) and followed to resolution as above. Patients should be seen at least 30 days after discontinuing study medication to collect and/or complete AE information.

# 5.9 Withdrawal from study

Patients are at any time free to withdraw from the study (study treatment and assessments), without prejudice to further clinical care (withdrawal of consent). Such patients should always be asked about the reason(s) and the presence of any adverse events. If possible, they will be seen and assessed by an investigator. Adverse events will be followed up (See Sections 6.4.9 and 6.4.10); questionnaires (e.g. for patient reported outcomes) and all study drugs should be returned by the patient.

Withdrawn patients will not be replaced.

Reasons for withdrawal from the study:

- Voluntary withdrawal by the patient who is at any time free to discontinue their participation in the study, without prejudice to further treatment\*
- Incorrectly enrolled patients i.e., the patient does not meet the required inclusion/exclusion criteria for the study this option is only applicable to patients not randomised into the study (i.e. screen failures identified prior to randomisation)
- Patient lost to follow-up
- Death

\*If a patient decides at any point in the trial that they do not wish to continue with the full study schedule of assessments but are still willing to provide important study information (e.g. disease recurrence information and/or survival status information) then the patient should continue in the study and information should continue to be collected in the eCRF. However, if a patient does not wish to have any further data collected, only then should they be considered as withdrawing consent from the study. To minimise the number of cases of early withdrawal the investigator should discuss the options with the patient to see if they would still be willing to provide

NCI Version Date: 05-06-2021 89(177) NSABP B-55/BIG 6-13

information on the important study endpoints (disease recurrence and overall survival), in which case they would remain in the study.

If a patient withdraws consent (i.e. nor further assessment or collection of their data), he/she should be specifically asked if they are also withdrawing consent to the use of any of their samples (tumour and blood) taken during the trial (see Sections 6.6, 6.7 and 6.8).

Data obtained prior to withdrawal of consent will be maintained in the clinical database and used in the study reporting.

#### 6. COLLECTION OF STUDY VARIABLES

# 6.1 Recording of data

# 6.1.1 Instructions for completion of B-55/6-13 forms and materials

Data form worksheets are available on the CTSU Member Web site, <a href="https://www.ctsu.org">https://www.ctsu.org</a>. A generic transmittal form can be created through the "Study Management" link located in Coordinator Online on the Members' Area of the NSABP Web site. Contact the Support @nrgoncology.org for an account to access the NSABP Web site.

#### 6.1.2 Instructions for submission of B-55/6-13 data, forms, and materials

• B-55/6-13 will use Medidata Rave for remote data capture of all data including routine adverse event reporting. The investigator will ensure that data are recorded on the eCRFs as specified in the study protocol and in accordance with the instructions provided. Query generation and resolution for B-55/6-13 are part of the Rave program. All queries will be issued and responded to electronically within Rave. Access to the trial in Rave is granted through the iMedidata application to all persons with the appropriate roles in Regulatory Support System (RSS). To access Rave via iMedidata, the site user must have an active CTEP-IAM account (check at < <a href="https://ctepcore.nci.nih.gov/iam">https://ctepcore.nci.nih.gov/iam</a>) and the appropriate Rave role (Rave CRA, Rave Read-Only, CRA [Lab Admin], SLA or Site Investigator) on either the LPO or participating organization roster at the enrolling site. To the hold Rave CRA role or CRA Lab Admin role, the user must hold a minimum of an AP registration type. To hold the Rave Site Investigator role, the individual must be registered as an NPIVR or IVR. Associates can hold read-only roles in Rave.

Upon initial site registration approval for the study in RSS, all persons with Rave roles assigned on the appropriate roster will be sent a study invitation e-mail from iMedidata. To accept the invitation, site users must log into the Select Login (<a href="https://login.imedidata.com/selectlogin">https://login.imedidata.com/selectlogin</a>) using their CTEP-IAM user name and password, and click on the "accept" link in the upper right-corner of the iMedidata page. Please note, site users will not be able to access the study in Rave until all required Medidata and study specific trainings are completed. Trainings will be in the form of electronic learnings (eLearnings), and can be accessed by clicking on the link in the upper right pane of the iMedidata screen.

Users that have not previously activated their iMedidata/Rave account at the time of initial site registration approval for the study in RSS will also receive a separate invitation from iMedidata to activate their account. Account activation instructions are located on the CTSU

NCI Version Date: 05-06-2021 90(177) NSABP B-55/BIG 6-13

website, Rave tab under the Rave resource materials (Medidata Account Activation and Study Invitation Acceptance). Additional information on iMedidata/Rave is available on the CTSU Members' website under the Rave tab at <a href="https://www.ctsu.org/RAVE/">https://www.ctsu.org/RAVE/</a> or by contacting the CTSU Help Desk at 1-888-823-5923 or by e-mail at <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>.

The investigator ensures the accuracy, completeness, and timeliness of the data recorded and of the provision of answers to data queries according to the Clinical Study Agreement.

The investigator will sign the completed eCRFs. A copy of the completed eCRFs will be archived at the study site.

Exceptions to submission of data through Medidata Rave are the signed and dated informed consent form, the BAHO questionnaire, and required source documents which should be faxed to the NRG Oncology SDMC according to the instructions on the form worksheet. When submission of supporting documentation to the NRG Oncology SDMC is required, fax to 412-622-2111. Remove patient names and identifiers such as social security number, address, telephone number, etc. from reports and supporting documentation. Do not include a cover sheet for faxed data.

# 6.1.3 Data monitoring for CTEP

This study will be monitored by the Clinical Data Update System (CDUS) Version 3.0. CTEP has assigned abbreviated CDUS reporting: no AE reporting (routine or expedited) is required via any of the CDUS mechanisms. Cumulative CDUS data will be submitted quarterly by the NRG Oncology SDMC to CTEP by electronic means. Reports are due January 31, April 30, July 31, and October 31.

Note: B-55/6-13 has been assigned to CDUS-Abbreviated reporting, no adverse event reporting (routine or expedited) is required to be reported via CDUS, but expedited adverse events are still required to be submitted via CTEP-AERS.

# 6.2 Study procedures

A schedule for the tests and evaluations to be conducted in this study is contained in this section and in <u>Table 1</u>, <u>Table 2</u>, and <u>Table 3</u>.

#### **6.2.1** Screening procedures

The following assessments, procedures, and data collection should be performed during screening as per <u>Figure 1</u> and <u>Table 1</u>.

- Provision of informed consent
- Assessment of eligibility against inclusion/exclusion criteria
- Date of birth
- Collect data on race and ethnicity
- Current and concomitant medications including previous cancer therapies

- Medical and surgical history including previous cancer and radiotherapy and history of blood transfusions in previous 120 days
- Family history of cancer
- Physical examination
- Vital signs (blood pressure and pulse; body temperature), body weight, height
- ECG (within 28 days prior to randomisation)
- Haematology/Clinical chemistry/Coagulation (see Section 6.4.11.2)/Urinalysis
- ECOG Performance Status
- If a patient with conservative surgery does not have a mammogram or breast MRI within 12 months prior to Screening PART 1, then this assessment must be performed prior to randomisation. Breast imaging should be performed on any remaining intact breast. Radiological tests to exclude a second primary breast cancer (either ipsilateral and/or contralateral) are mandatory before enrolment (within 12 months prior to Screening PART 1) for patients with any remaining intact breast tissue. The preferred tests are mammograms or MRI (MRI preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion.
- Pregnancy tests on serum or urine samples will be performed for women of childbearing potential within 28 days prior to randomisation and on Day 1 of the study prior to commencing treatment.
- CPS+EG score (Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS)) for the non-pCR patients who received prior neoadjuvant chemotherapy (Mittendorf et al 2011; Jeruss et al 2008). Instructions on how to calculate the CPS&EG score are provided in Appendix H.
- Patient Reported Outcomes and Quality of life questionnaire: FACIT-Fatigue and EORTC QLQ-C30 will be collected prior to randomisation once eligibility is confirmed.
- Germline BRCA1/2 mutation status determination
  - All patients must have a known deleterious or suspected deleterious germline BRCA mutation to be randomised; this may have been determined by local genetic testing prior to enrolment into the study or may be assessed as part of the enrolment procedure for the study which requires a central laboratory test at Myriad Genetics, Inc.

NCI Version Date: 05-06-2021 92(177) NSABP B-55/BIG 6-13

- Two blood samples are mandated for all patients, one sample will be used to test for BRCA mutations using the current commercial Myriad BRCAnalysis test, and the second sample is required for a bridging study to validate the companion diagnostic test for olaparib.
- O Patients with unknown *BRCA* status must have a central test performed by Myriad prior to randomisation into the study. Patients will need to have met the locally agreed guidelines for *BRCA* testing with genetic counselling arranged as appropriate. When the result from the Myriad test indicates the patient does have a deleterious or suspected deleterious *BRCA* mutation, and the patient meets all other eligibility criteria, the patient can be randomised into the study. Specimen collection and results disclosure to the potential subject will be conducted using local ethical procedures.
- o It is recommended that, where required, the Myriad gBRCA test is undertaken during adjuvant or neoadjuvant chemotherapy to allow time for necessary counselling and for the return and discussion of the test result.
- o Patients with known deleterious or suspected deleterious *BRCA* mutation/s prior to enrolment into the study can be randomised into the study based on this local result provided they meet all other eligibility criteria. The specific *BRCA1/2* mutation must be reported in the clinical database by selecting the appropriate value from the drop down menu. At screening, reconfirmation of the *BRCA* mutation from a blood sample will be undertaken by a central laboratory (Myriad Genetics, Inc.). Should the result from the central Myriad test indicate that the patient does not have a deleterious or suspected deleterious *BRCA* mutation, this information will be available to the study investigator and the decision as to whether or not the patient continues study treatment should be made between the patient and study investigator.
- o If the discordance is based on the absence of the alteration identified in the local laboratory by the central laboratory, then analysis of a second specimen, collected independently from the patient and sent to Myriad Genetics, Inc. for re-analysis of the presence or absence of the mutation specified in the original test or otherwise as discussed with Myriad laboratory staff, may be performed under the protocol, to eliminate sample mislabelling and similar errors. These errors are expected to be uncommon. If the discordance is based on interpretation of the pathogenicity of an alteration identified by both laboratories (i.e., Myriad classifies the alteration as neither deleterious nor suspected deleterious), a repeat test will not be indicated. The OlympiA trial Genetic Advisory Committee can be consulted if needed.

See Section 6.6.2 for gBRCA Myriad samples collection.

• Adverse events must be captured from time of main consent. Any medical condition (new or worsening of a pre-existing condition) that occurs post Screening PART 2 and is continuing at randomisation should be recorded in Medical History in the eCRF as a medical condition current at randomisation. If the condition worsens post randomisation, this should be recorded as an AE/SAE in the eCRF with start date as the date the grade worsened and the new grade should be reported on the AE form. The AE/SAE would be

NCI Version Date: 05-06-2021 93(177) NSABP B-55/BIG 6-13

considered to have resolved when it resolves to the baseline grade, not to zero. Any medical condition considered of clinical relevance (new or worsening of a pre-existing condition) that occurs post consent for PART 2 and resolves prior to randomisation should also be recorded as medical history. In Screening PART 1 of the study only SAEs related to study mandated procedures (i.e., blood draw) will be collected. In Screening Part 2 all SAEs will be collected. For the patients who experienced an SAE in either Screening PART 1 or PART 2 that were eventually randomised, the SAE should be reported in the eCRF retrospectively in addition to paper reporting as described in Section 6.4.9 and Section 6.4.10.

- Check availability of an archival paraffin embedded tumour tissue sample (see <u>Section 6.6.3</u>). (The sample will only be submitted to the study bio-repository once the patient has been randomised.)
- Check availability of an archival paraffin embedded post neoadjuvant tumour tissue sample (see <u>Section 6.6.4</u>). (The sample is required from neoadjuvant patients only and will only be sent to the study bio-repository once the patient has been randomised.)

The Principal Investigator/Sub-Investigator should adhere to the study plan, procedures and perform tests/observations in accordance with the protocol.

#### 6.2.2 On-treatment assessments

Patients will attend the clinic on day 1 (1st day of treatment) and, following the commencement of 300 mg b.i.d twice daily dosing, every 2 weeks during the first month, every 4 weeks for the following 5 months and 3 monthly for the remaining 6 months of study treatment plus 30 days after its discontinuation.

The following assessments will be performed at time points specified in the study schedule (see Section 3.1, Table 1 and Table 2):

- Physical examination (data need not be entered in the eCRF, however any clinically significant changes from baseline must be reported as an AE or an event) e.g. any signs of recurrence of disease should be reported
- ECOG performance status: if assessed within 7 days of randomisation, it should not be assessed again at day 1 of study treatment
- Vital signs (blood pressure and pulse rate, body temperature, body weight): if assessed within 7 days of randomisation, are not required to be assessed again at day 1 of 1st day of study treatment
- Haematology and clinical chemistry: Safety blood samples do not need to be repeated on Day 1 of study treatment if there have been separate assessments within 7 days before randomisation and at least 3 weeks after last dose of chemotherapy, unless the investigator believes that it is likely to have changed significantly

NCI Version Date: 05-06-2021 94(177) NSABP B-55/BIG 6-13

- Race and ethnicity unless collection of this data is not allowed by local regulation
- Pregnancy tests on serum or urine samples will be performed for women of childbearing potential. If the test is positive the patient is ineligible/must be discontinued from study treatment immediately.
- AE and concomitant medications (including any blood transfusions) at every visit
- Patient Reported Outcomes and Quality of life questionnaire: FACIT-Fatigue and EORTC QLQ-C30 will be collected at 6 months, 12 months, 18 months and 24 months



- Optional pharmacokinetic samples will be obtained from consenting patients on day 29 (see <u>Section 6.8</u>). PK sampling not being done in the US.
- Optional tumour biopsy at disease recurrence (Section 6.6.5)
- Mandatory blood sample for biomarker analysis (e.g. cfDNA) on day 1 prior to first dose of study treatment, 30 days post study treatment and disease recurrence (Section 6.6.6)
- Radiological tests to exclude a second primary breast cancer (ipsilateral and/or contralateral) are mandatory during study participation (starting at week 24 and yearly thereafter) for patients with any remaining intact breast tissue. The preferred tests are mammogram or MRI (MRI preferred for patients below 50 years of age). For patients who underwent a bilateral mastectomy, with no remaining breast tissue, a physical examination is sufficient and radiological tests are not mandatory. For patients who underwent a bilateral mastectomy, as well as for male patients, clinical exam may be supplemented by ultrasound exams at investigator's discretion.
- Dispensing of and return of unused study treatment

Within this study, patients will not be provided olaparib post discontinuation of study treatment. Patients and investigators will not be unblinded to study treatment prior to the final overall survival (OS) analysis.

#### 6.2.3 Efficacy follow-up assessments

Assessments for disease recurrence, new cancers and overall survival will be performed based on signs and symptoms, clinical assessment (i.e. physical exam), mammograms and/or breast MRI and vital status.

Following randomisation, during the first 2 years patients will be assessed for disease recurrence and new cancers every 3 months. During years 3, 4 and 5 patients will be assessed every

6 months and then annually until approximately 10 years from randomisation if an IDFS endpoint due to a distant breast cancer relapse has not been met.

Mammograms and/or MRI (MRI preferred for patients younger than 50 years) (ipsilateral and/or contralateral) will be performed annually in patients with retained breast tissue beginning 6 months after the first day of treatment for approximately 10 years if an IDFS endpoint due to a distant breast cancer relapse has not been met.

Once a patient has received clinical follow-up for efficacy for approximately 10 years, or an IDFS endpoint due to a distant breast cancer relapse has been met, the patient will then enter the annual survival follow-up phase of the study. During the survival follow-up phase, no clinic visits will be required; information may be collected via telephone, medical records or death registries. Vital status information, as well as other information specified in footnote g of <u>Table</u> 2, will be collected until 10 years after the last patient is randomised.

In addition to disease status and vital status, information on first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time, including those received during the survival follow-up phase, will be collected. Information on endocrine therapies should be collected and recorded in the eCRF until IDFS endpoint is met due to breast cancer related distant relapse. The therapy type and start and stop dates of therapy will be collected.

# 6.2.4 Safety follow-up assessments 30 days after last dose of olaparib/placebo

A follow-up visit should be conducted 30 days after the last dose of olaparib/placebo. Any serious and/or non-serious AEs ongoing at the time of discontinuation of study treatment or which have occurred during the defined 30-day follow-up period must be followed-up (in accordance with Section 6.4.9). Appropriate safety evaluations should be repeated and/or additional tests performed at any time when clinically indicated, or at the discretion of the investigator, until resolution, unless, in the investigator's opinion, the condition is unlikely to resolve due to the patient's underlying disease. If the patient is lost to follow-up, then this should be noted in the eCRF. The assessments to be carried out at the 30-day follow up visit are detailed in the study schedule (Table 2).

See Section 6.4.9 for details of long term safety collection.

# 6.2.5 Patient management post-primary analysis

The data cut off (DCO) for the primary analysis for IDFS will occur once 330 IDFS events have been reported. Once this data is fully validated the primary analysis will be conducted and reported.

At the time of the DCO for the primary analysis patients will continue in the study as per the protocol following the outlined study plan assessments. Patients who have completed treatment and all relevant safety assessments will continue to have regular efficacy assessments as detailed in the study plan. All ongoing patients will continue to be followed for recurrence, new cancers and overall survival irrespective of treatment status.

NCI Version Date: 05-06-2021 96(177) NSABP B-55/BIG 6-13

It is anticipated that further analysis of the efficacy data, particularly the secondary endpoints, will be conducted with more mature follow up. Any further available safety data will also be reported.

#### 6.2.6 Patient management post-final analysis

Study follow up will continue until approximately 10 years after the last patient is randomised. After this time no further data collection is anticipated.

Patient management post the final analysis will be according to local clinical practice. All patients will have completed study treatment by the time of the final analysis.

# 6.3 Efficacy

#### **6.3.1** Tumour evaluation

All treatment decisions and analysis for this study will be based on investigator evaluation of assessments. Following randomisation, all patients will be assessed regularly for signs, symptoms and evidence of disease recurrence by reviewing medical history, performing physical examination and mammogram and/or breast MRI (MRI preferred for patients younger than 50 years). See <u>Table 2</u> and <u>Table 3</u>. Efficacy assessments (medical history and physical examination) will be performed on a 3 monthly basis during the first 2 years, followed by 6 monthly assessments for years 3, 4 and 5 and annually thereafter. All patients will have mammogram and/or breast MRI (ipsilateral and/or contralateral) annually for approximately 10 years beginning 6 months after day 1. Evidence of disease recurrence or new primary cancer will require histopathological and/or radiological confirmation.

Patients will be regularly assessed, through clinical visits, for recurrence (local and distant) and new cancers for approximate 10 years follow-up regardless of whether they have discontinued study treatment or started any subsequent anti-cancer therapies. Following completion of approximately 10 years' clinical follow-up assessments, patients will enter a survival follow-up phase, which will continue until 10 years after the last patient is randomised. During the survival contact period information on any known subsequent sites of metastases, new cancers and further subsequent therapies (information on first line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time) will be captured as well as vital status. Study visits are not required during the survival follow-up phases; contact may be made via telephone, medical records or death registries once per year.

Loco-regional recurrence of the disease (ipsilateral or regional invasive breast cancer) should be cytologically/histologically confirmed. Imaging to assess for distant metastatic disease or any other area as clinically indicated should be performed at the time of local recurrence to ensure that any further spread of the disease is detected. Isolated loco-regional recurrence should be managed with curative intent when possible. Suspected distant recurrence should be confirmed by radiological examination and every attempt made to obtain histopathological confirmation when a metastatic lesion is easily accessible for biopsy. Invasive contralateral breast cancer or invasive non-breast secondary primary cancer should be confirmed by histopathology.

NCI Version Date: 05-06-2021 97(177) NSABP B-55/BIG 6-13

Patients who develop loco-regional recurrence should discontinue study treatment (if within the study treatment period) but will continue to be followed for distant recurrence (including subsequent sites of metastases) and all new cancers (local, regional, second primary malignancy or contralateral breast cancer), subsequent therapies and survival as per study schedule. The first EVENT (local, regional or distant recurrence, second primary malignancy or contralateral breast cancer) should be recorded in the eCRF. The following additional information should also be recorded in the eCRF along with the results of the confirmatory tests.

- First distant relapse (if not the first EVENT);
- CNS metastases, that should always be reported regardless of any prior recurrences;
- Local regional relapses, occurring after the first event;
- Contralateral breast cancer, at any time;
- Any second primary malignancies, at any time.

Patients who develop distant recurrence should discontinue study treatment (if within the study treatment period) but will continue to be followed for development of additional sites of metastatic disease, new cancers, subsequent therapies and survival as per the survival follow-up schedule.

Disease recurrence or new cancers should be reported in the eCRF as soon as possible after they are discovered. This includes events diagnosed during study visits but also any event diagnosed during non-study visits.

Once known, death information should also be recorded in the eCRF as soon as possible.

# 6.4 Safety

The Principal Investigator is responsible for ensuring that all staff involved in the study is familiar with the content of this section.

# 6.4.1 Investigational agents

The investigational agent administered in B-55/6-13 is olaparib, which is being made available under an IND sponsored by NRG Oncology, Inc. Expectedness of adverse events is based on the current IB.

#### 6.4.2 Commercial agents

There are no commercial supply agents in B-55/6-13.

# 6.4.3 Double-blind study drug

This is a double-blind study and includes an investigational agent with placebo. When an AE occurs that is expected for the investigational agent, the AE should be considered expected for the blinded study therapy. Conversely, when an adverse event occurs that is not listed for the investigational agent, the AE should be considered to be unexpected for the blinded therapy.

#### 6.4.4 Adverse event characteristics

CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. CTCAE version 5.0 is being utilized for SAE reporting as of April 1, 2018. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0 and the CTCAE version 5.0. A copy of the CTCAE version 4.0 and CTCAE version 5.0 can be downloaded from the CTEP Web site (http://ctep.cancer.gov).

# 6.4.5 Definition of adverse events (AE)

An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g. nausea, chest pain), signs (e.g. tachycardia, enlarged liver) or the abnormal results of an investigation (e.g. laboratory findings, electrocardiogram).

The term AE is used to include both serious and non-serious AEs.

# 6.4.6 Definitions of serious adverse event (SAE)

A serious adverse event is an AE occurring during any study phase (i.e. from the time a patient signs a study specific consent form, treatment, and follow-up), that fulfils one or more of the following criteria:

- Results in death
- Is immediately life-threatening
- Requires in-patient hospitalisation or prolongation of existing hospitalisation
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital abnormality or birth defect
- Is an important medical event that may jeopardise the patient or may require medical intervention to prevent one of the outcomes listed above.

For further guidance on the definition of an SAE, see <u>Appendix A</u> to the Clinical Study Protocol.

#### 6.4.7 Common adverse events associated with olaparib

Following is a list of common AEs associated with olaparib. Refer to the current IB for complete toxicity information.

- Blood and Lymphatic System Disorders Anemia
- Gastrointestinal Disorders Abdominal pain; Bloating; Diarrhea; Dyspepsia; Mucositis oral; Nausea; Vomiting
- General Disorders and Administration Site Conditions Edema limbs; Fatigue, Fever
- Immune System Disorders Allergic reaction

- *Investigations* Creatinine increased; Investigation Other, mean corpuscular volume; Lymphocyte count decreased; Platelet count decreased
- Metabolism and Nutrition Disorders Anorexia
- Neoplasms benign, malignant and unspecified (incl cysts and polyps Leukemia secondary to oncology chemotherapy; Myelodysplastic syndrome; Treatment related secondary malignancy
- Nervous System Disorders Dizziness; Dysgeusia; Headache
- Respiratory, Thoracic, and Mediastinal Disorders Cough; Dyspnea; Pneumonitis
- Skin and Subcutaneous Tissue Disorders Dermatitis; Rash maculo-papular

# **6.4.8** Expedited reporting of adverse events

NRG Oncology follows procedures for centralized reporting of adverse events, which requires that adverse events/serious adverse events be reported to the NRG Oncology SDMC. NRG Oncology forwards reports to the appropriate regulatory agencies and the pharmaceutical company involved in the trial.

All serious adverse events that meet expedited reporting criteria defined in <u>Table 11</u> will be reported via the CTEP Adverse Event Reporting System, CTEP-AERS, accessed via the CTEP web site, <a href="https://eapps-ctep.nci.nih.gov/ctepaers">https://eapps-ctep.nci.nih.gov/ctepaers</a>. NRG Oncology is identified in CTEP-AERS as the Lead Group for CTEP-AERS reporting.

Submitting a report via CTEP-AERS serves as notification to the NRG Oncology Statistics and Data Management Center (SDMC) and satisfies NRG Oncology requirements for expedited adverse event reporting.

In the rare event when Internet connectivity is disrupted, a 24-hour notification is to be made to the NRG Oncology SDMC by telephone at 412-383-2557. An electronic report must be submitted immediately upon re-establishment of the Internet connection.

For questions concerning expedited AE reporting, contact the B-55/6-13 AE reporting nurse (see Information Resources).

# **6.4.8.1** Expedited reporting methods

- Per CTEP NCI Guidelines for Adverse Events Reporting Requirements, a CTEP-AERS
   24-Hour Notification must be submitted to the NCI within 24 hours of learning of the adverse event. Each CTEP-AERS 24-hour notification must be followed by a CTEP-AERS
   3 Calendar Day Report (see Table 11).
- CTEP-AERS 3 Calendar Day Report requires that a complete report is electronically submitted to the NRG Oncology Lead Group within 3 calendar days of submission of the CTEP-AERS 24-hour notification (see Table 11).
- CTEP-AERS 5 Calendar Day Report requires that a complete report is electronically submitted to the NRG Oncology Lead Group within 5 calendar days of learning of the AE (see Table 11).
- Reports submitted via CTEP-AERS 24-hour notification are available for review by both the NCI and NRG Oncology after submission. All other CTEP-AERS reports are first sent to the NRG Oncology Lead Group and then are forwarded to the NCI. The timelines in

NCI Version Date: 05-06-2021 100(177) NSABP B-55/BIG 6-13

<u>Table 11</u> have been set so that the information can be forwarded to the NCI in a timely manner per the NCI's/CTEP's guidelines.

• Supporting documentation is requested by the IND sponsor for this study (NRG Oncology) as needed to complete adverse event review. All CTEP-AERS documentation is faxed to NRG Oncology SDMC at 412-622-2113. When submitting supporting source documentation, remove all identifiers and include the protocol number, patient ID number, and CTEP-AERS ticket number on each page.

# 6.4.8.2 Protocol-specific expedited reporting requirements

**Protocol-specific expedited reporting requirements**: For this study, the following adverse events require expedited reporting via CTEP-AERS to the NRG Oncology Lead Group **within 5 calendar days** (or sooner if required based on other <u>Table 11</u> instructions) of learning of the event:

Expedited reporting via CTEP-AERS is required for the following from the first dose of study therapy until the end of the patient's follow-up irrespective of the timing of the event in relation to study therapy):

- Leukemia secondary to oncology chemotherapy (e.g., acute myelocytic leukemia [AML])
- Myelodysplastic syndrome (MDS)
- Second primary malignancy
- Pneumonitis

Supporting documentation, including pathology and cytogenetics reports which confirm the second malignancy, must be faxed to the NRG Oncology SDMC expedited fax at 412-622-2113. Each page of supporting documentation must include the NCI protocol number, the CTEP-AERS ticket number, and the protocol-specific Patient ID number provided during trial registration.

Any second malignancy (including AML/MDS) should also be reported within the B-55/6-13 Follow-up folder in Medidata Rave. Fax supporting documentation that confirms the secondary malignancy diagnosis with the transmittal form to 412-622-2111.

NCI Version Date: 05-06-2021 101(177) NSABP B-55/BIG 6-13

Table 11 Late Phase 2 and Phase 3 Studies: Expedited reporting requirements for adverse events that occur on studies under an IND within 30 days of the last administration of the investigational agent (olaparib/placebo)<sup>1</sup>

# FDA REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS (21 CFR Part 312)

**NOTE:** Investigators <u>MUST</u> immediately report to the sponsor (NRG Oncology) <u>ANY</u> Serious Adverse Events, whether or not they are considered related to the investigational agent (21 CFR 312.64)

An adverse event is considered serious if it results in **ANY** of the following outcomes:

- 1) Death
- 2) A life-threatening adverse event
- 3) An adverse event that results in inpatient hospitalization or prolongation of existing hospitalization for ≥ 24 hours
- 4) A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5) A congenital anomaly/birth defect
- 6) Important Medical Events (IME) that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (FDA, 21 CFR 312.32; ICH E2A and ICH E6).

<u>ALL SERIOUS</u> adverse events that meet the above criteria <u>MUST</u> be immediately reported to the NCI and NRG Oncology via CTEP-AERS within the timeframes detailed in the table below.

| Hospitalization | Grade 1<br>Timeframes | Grade 2<br>Timeframes | Grade 3<br>Timeframes | Grade 4 & 5<br>Timeframes |
|---|---|---|---|---|
| Resulting in<br>Hospitalization<br>≥ 24 hrs | 5 Calendar Days | | | 24-Hour, |
| Not resulting in<br>Hospitalization<br>≥ 24 hrs | Not required | | 5 Calendar Days | 3 Calendar Days |

NOTE: See <u>Section</u> <u>6.4.8.2</u> for protocol-specific expedited reporting requirements and exceptions. Expedited AE reporting timelines are defined as:

- "24-Hour, 3 Calendar Days" The AE must initially be reported via CTEP-AERS within 24 hours
  of learning of the AE, followed by a complete expedited report submitted to the NRG Oncology
  Lead Group within 3 calendar days of the initial 24-hour report.
- "5 Calendar Days" A complete expedited report on the AE must be submitted within 5 calendar days of learning of the AE.

1Serious adverse events that occur more than 30 days after the last administration of investigational agent and have an attribution of possible, probable, or definite require reporting as follows:

Expedited 24-hour notification followed by complete report with 3 calendar days for:

• All Grade 4 and Grade 5 AEs

# Expedited 5 calendar days reports for:

- Grade 2 adverse events resulting in hospitalization or prolongation of hospitalization
- Grade 3 adverse events Effective Date: May 5, 2011

NCI Version Date: 05-06-2021 102(177) NSABP B-55/BIG 6-13

# 6.4.9 Recording of adverse events

# Time period for collection of adverse events

Adverse events will be collected from time of signature of main informed consent\* throughout the treatment period up to and including the 30-day follow-up period (see Section 6.2.4). All ongoing and any new AEs/SAEs identified during the 30 calendar day follow-up period after the last dose of study medication must be followed to resolution unless the event is considered by the investigator to be unlikely to resolve, or the patient is lost to follow-up or in survival follow-up. AstraZeneca retains the right to request additional information for any patient with ongoing AE(s)/SAE(s) at the end of the study, if judged necessary. Any medical condition (new or worsening of a pre-existing condition) that occurs post Screening PART 2 and is continuing at randomisation should be recorded in medical history in the eCRF as a medical condition current at randomisation. If the condition worsens post randomisation, this should be recorded as an AE/SAE in the eCRF with start date as the date the grade worsened and the new grade should be reported on the AE form. The AE/SAE would be considered to have resolved when it resolves to the baseline grade, not to zero. Any medical condition considered of clinical relevance (new or worsening of a pre-existing condition) that occurs post consent for PART 2 and resolves prior to randomisation should also be recorded as medical history. Any AE happening from randomisation to the 30-day follow-up period should be reported on the AE form in the eCRF. If an Investigator learns of any SAEs, including death, at any time after a patient has completed the 30 days post treatment follow-up period, and he/she considers there is a reasonable possibility that the event is causally related to the study treatment, the investigator should report the SAE via CTEP-AERS (see Sections 6.4.9 and 6.4.10 and Table 11).

Any case of MDS/AML or new second primary malignancy occurring at any time from signature of informed consent for the entire participation of the patient in the study including the follow-up period should be reported as a SAE via CTEP-AERS, regardless of the investigator's assessment of causality, knowledge of the treatment arm, and irrespective of the timing of the event in relation to study therapy. All non-melanoma invasive skin cancers and all carcinoma in situ cases need to be reported as a non-serious AE unless at least one of the seriousness criteria is met and then it must be reported as an SAE (see Section 6.4.6). If a patient develops MDS/AML, full diagnostic details and classification should be provided e.g. bone marrow and cytogenetic analysis reports, see Sections 5.5.12.4 and 6.4.11.5. A questionnaire will be sent to any investigator reporting MDS/AML or new primary malignancy so that relevant details can be reported.

\*In Screening PART 1 of the study only SAEs related to study mandated procedures (i.e. blood draw) will be collected. In Screening PART 2 all SAEs will be collected (see <u>Table 1</u>). For the patients who experienced an SAE in either Screening PART 1 or PART 2 that were eventually randomised, the SAE should be reported in the eCRF retrospectively in addition to reporting the SAE via CTEP-AERS as described in Sections 6.4.9 and 6.4.10 and Table 11)

NCI Version Date: 05-06-2021 103(177) NSABP B-55/BIG 6-13

#### Adverse events after the 30-day follow up period

For pharmacovigilance purposes and characterisation, any SAE of MDS/AML, new second primary malignancy (with the exception of non-melanoma skin cancers and carcinoma in situ), or pneumonitis occurring after the 30-day follow up period should be reported as a SAE via CTEP-AERS regardless of investigator's assessment of causality, knowledge of the treatment arm, and irrespective of the timing of the event in relation to study therapy (see Section 6.4.8.2).

At any time after a patient has completed the study, if an investigator learns of any SAE including sudden death of unknown cause, and he/she considers there is a reasonable possibility that the event is causally related to the investigational product, the SAE should be reported via CTEP-AERS.

Otherwise, after study treatment completion (i.e. after any scheduled post treatment follow-up period has ended) there is no obligation to actively report information on new AEs or SAEs occurring in study patients. This includes new AEs/SAEs in patients still being followed up for survival but who have completed the post treatment follow up period (30 days).

#### Follow-up of unresolved adverse events

Any SAEs or non-serious adverse event that is still ongoing during the 30-day follow-up visit must be followed up to resolution unless the event is considered by the investigator to be unlikely to resolve, or the patient is lost to follow-up. AstraZeneca may request additional information for any patient with ongoing AE(s)/SAE(s) at the end of the study, if necessary.

# Reporting routine adverse events through Medidata Rave

- Reporting of routine adverse events is done through Medidata Rave.
- All ≥ grade 1 adverse events that occurred during study therapy must be reported on the B-55/6-13 Adverse Event forms (the Listed Adverse Event form or the Other Adverse Event form) through Medidata Rave, regardless of whether these adverse events are expected or unexpected.
- All adverse events reported via CTEP-AERS must also be reported on the B-55/6-13 Adverse Event forms through Medidata Rave.
- Supporting documentation for each AE reported on either of the B-55/6-13 Adverse Event forms through Medidata Rave must be maintained in the patient's research record. When submission of supporting documentation to the NRG Oncology SDMC is required, fax with a transmittal form to 412-622-2111. Remove patient names and identifiers such as social security number, address, telephone number, etc., from reports and supporting documentation.

#### **Variables**

The following variables will be collected for each AE;

- AE description (verbatim)
- The dates when the AE started and stopped

NCI Version Date: 05-06-2021 104(177) NSABP B-55/BIG 6-13

- CTCAE grade and changes in CTCAE grade
- Whether the AE is serious or not
- Investigator causality rating against the study treatment (yes or no)
- Action taken with regard to study treatment
- Outcome.

In addition, the following variables will be collected for SAEs:

- Date that the AE met criteria for serious AE
- Date Investigator became aware of serious AE
- Reason for AE being considered serious
- Date of hospitalisation
- Date of discharge
- Probable cause of death
- Date of death
- Autopsy performed
- Causality assessment in relation to Study treatment or procedure(s)
- Causality assessment in relation to Other medication
- Description of AE.

#### **Severity of AE**

For each episode of an adverse event, all changes to the CTCAE grade attained as well as the highest attained CTC grade should be reported.

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria in <u>Section 6.4.6</u>. An AE of severe intensity should not necessarily be considered serious. For example, nausea that persists for several hours may be considered severe nausea, but not an SAE. On the other hand, a stroke that results in only a limited degree of disability may be considered a mild stroke but would be an SAE.

The grading scales found in the National Cancer Institute (NCI) CTCAE version 4.0 will be utilised for all events with an assigned CTCAE grading. For those events which do not fall under any of the CTCAE defined categories, the investigator should assess them as mild, moderate severe, or life-threatening, or, if the patient dies, as an event leading to the patient's death.

NCI Version Date: 05-06-2021 105(177) NSABP B-55/BIG 6-13

A copy of the CTCAE version 4.0 can be downloaded from the NCI Cancer Therapy Evaluation Program website <a href="http://ctep.cancer.gov/">http://ctep.cancer.gov/</a>.

# **Causality collection**

The Investigator will assess causal relationship between study treatment and each Adverse Event, and answer 'yes' or 'no' to the question 'Do you consider that there is a reasonable possibility that the event may have been caused by the study treatment?'

For SAEs causal relationship will also be assessed for other medication and study procedures. Note that for SAEs that could be associated with any study procedure the causal relationship is implied as 'yes'.

A guide to the interpretation of the causality question is found in <u>Appendix A</u> to the Clinical Study Protocol.

# Adverse events based on signs and symptoms

All AEs spontaneously reported by the patient or reported in response to the open question from the study personnel: 'Have you had any health problems since the previous visit/you were last asked?', or revealed by observation will be collected and recorded in the eCRF and submitted. When collecting AEs, the recording of diagnoses is preferred (when possible) rather than recording a list of signs and symptoms. However, if a diagnosis is known and there are other signs or symptoms that are not generally part of the diagnosis, the diagnosis and each sign or symptom will be recorded separately.

#### Adverse events based on examinations and tests

The reporting of laboratory/vital signs/ECG abnormality as an AE should be avoided unless one of the following is met:

- Any criterion for an SAE is fulfilled
- Causes study treatment discontinuation
- Causes study treatment interruption
- Causes study treatment dose reduction
- The investigator believes that the abnormality should be reported as an AE

If deterioration in a laboratory value/vital sign is associated with clinical signs and symptoms, the sign or symptom will be reported and submitted as an AE and the associated laboratory result/vital sign will be considered as additional information. Wherever possible the reporting investigator uses the clinical, rather than the laboratory term (e.g. anaemia versus low haemoglobin value). In the absence of clinical signs or symptoms, clinically relevant deteriorations in non-mandated parameters should be reported and submitted as AE(s).

NCI Version Date: 05-06-2021 106(177) NSABP B-55/BIG 6-13

Deterioration of a laboratory value, which is unequivocally due to disease recurrence, should not be reported as an AE/SAE.

Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the baseline assessment will be reported and submitted as an AE.

**NB.** Cases where a patient shows an AST or ALT  $\ge 3x$ ULN or total bilirubin  $\ge 2x$ ULN may need to be reported as SAEs, please refer to <u>Appendix D</u> 'Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law', for further instructions.

#### Disease recurrence

The development of loco-regional recurrence or distant metastasis to the primary cancer under study should be considered as disease progression and not an AE. Events, which are unequivocally due to disease recurrence, should not be reported as an AE during the study.

Report breast cancer recurrence within the B-55/6-13 Follow-up folder in Medidata Rave. Fax supporting documentation that confirms the breast cancer recurrence with the transmittal form to 412-622-2111.

# New primary cancers (second malignancy)

The development of a new primary cancer (second malignancy) should be reported as a SAE. New primary cancers are those that are not the primary reason for the administration of the study treatment and have developed after the inclusion of the patient into the study. They do not include metastases of the original cancer. Symptoms of metastasis or the metastasis itself should not be reported as an AE/SAE, as they are considered to be disease recurrence. New primary cancers are considered as IDFS events and must also be reported on the endpoint CRF. Patients with new primary cancers that can be adequately treated with surgery only and which do not require any additional (neo)adjuvant treatment of any kind can continue to receive investigational product and be followed for secondary endpoints. Rules regarding temporary interruption due to surgery apply (see Section 5.5.12.7). Patients with new primary cancers which require (neo)adjuvant treatment of any kind for appropriate management must be discontinued from study treatment.

#### **Deaths**

All deaths that occur during the study (see Section 6.4.9) must be reported as follows:

- Death that is clearly the result of breast cancer recurrence or progression should be reported in the DEATH eCRF but should not be reported as an SAE
- Where death that occur within 30 days of the last dose of study treatment is not due (or not clearly due) to breast cancer recurrence or progression of the disease under study, the cause of death must be reported via CTEP-AERS as a SAE within 24 hours (see Section 6.4.10 for further details). The report should contain a comment regarding the co-involvement of progression of disease, if appropriate, and should assign main and contributory causes of death. This information should be captured in the relevant eCRF.

NCI Version Date: 05-06-2021 107(177) NSABP B-55/BIG 6-13

- Deaths with an unknown cause that occur within 30 days of the last dose of study treatment must be reported via CTEP-AERS. A post mortem maybe helpful in the assessment of the cause of death, and if performed a copy of the post-mortem results should be forwarded to the NRG Oncology SDMC within the usual timeframes.
- A copy of the death certificate should be forwarded to the NRG Oncology SDMC if it is readily available or if it contains important cause-of-death information that is not documented elsewhere.
- Please submit the last clinical/office note made before the death or the investigator's note summarizing events resulting in death.

# Olaparib adverse events of special interest

Adverse events of special interest (AESI) are events of scientific and medical interest specific to the further understanding of olaparib's safety profile and require close monitoring and reported via CTEP-AERS. Adverse Events of Special Interest for olaparib are MDS/AML, new second primary malignancy (other than MDS/AML) and pneumonitis.

A questionnaire will be sent to any investigator reporting an AESI as an aid to provide further detailed information on the event. During the study there may be other events identified as AESIs that require the use of a questionnaire to help characterise the event and gain a better understanding regarding the relationship between the event and study treatment.

# 6.4.10 Reporting of serious adverse events

All SAEs have to be reported, whether or not considered causally related to the study treatment or to the study procedure(s). All SAEs will be reported via CTEP-AERS and Medidata Rave (see Section 6.4.8, Section 6.4.9, and Table 11).

The NRG Oncology site AE reporter works with the investigator to ensure that all the necessary information is provided within one calendar day of initial receipt for fatal and life threatening events and within five calendar days of initial receipt for all other SAEs.

If CTEP-AERS is not available, refer to <u>Section</u> <u>6.4.8</u> for reporting instructions.

# 6.4.11 Laboratory safety assessment

Blood and urine samples for determination of clinical chemistry, haematology, coagulation, and urinalysis will be taken at the times indicated in the Study Schedule (see <u>Table 1</u> and <u>Table 2</u>).

These tests will be performed by the hospital's local laboratory. Additional analyses may be performed if clinically indicated.

Any clinically significant abnormal laboratory values should be repeated as clinically indicated and recorded on the eCRF.

The following laboratory variables will be measured:

NCI Version Date: 05-06-2021 108(177) NSABP B-55/BIG 6-13

# 6.4.11.1 Full haematology assessments for safety

- haemoglobin
- red blood cells [RBC]
- platelets
- mean cell volume [MCV]
- mean cell haemoglobin concentration [MCHC]
- mean cell haemoglobin [MCH]
- white blood cells [WBC]
- absolute differential white cell count
  - (neutrophils, lymphocytes, monocytes, eosinophils and basophils) and absolute neutrophil count or segmented neutrophil count and Band forms should be performed at each visit and when clinically indicated. If absolute differentials not available please provide % differentials

# 6.4.11.2 Coagulation

- activated partial thromboplastin time (APTT) will be performed at baseline and if clinically indicated
- international normalised ratio (INR) will be performed at baseline and if clinically indicated unless the patient is receiving warfarin. Patients taking warfarin may participate in this study; however, it is recommended that prothrombin time (INR and APTT) be monitored carefully at least once per week for the first month, then monthly if the INR is stable

#### 6.4.11.3 Clinical chemistry assessments for safety

- sodium
- potassium
- calcium
- creatinine
- total bilirubin
- alkaline phosphatase [ALP]

NCI Version Date: 05-06-2021 109(177) NSABP B-55/BIG 6-13

- aspartate transaminase [AST]
- alanine transaminase [ALT]
- urea or blood urea nitrogen [BUN]
- total protein
- albumin

**NB.** If a patient has AST or ALT  $\geq$  3xULN or total bilirubin  $\geq$  2xULN please refer to <u>Appendix</u>  $\underline{D}$  'Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law', for further instructions.

For blood volume see Section 7.1.

#### **6.4.11.4** Urinalysis

Urinalysis by dipstick should be performed at baseline and then only if clinically indicated. Microscopic analysis should be performed by the hospital's local laboratory if required.

# 6.4.11.5 Bone marrow or blood cytogenetic samples

Bone marrow or blood cytogenetic samples may be collected for patients with prolonged haematological toxicities as defined in <u>Section 5.5.12.4</u>.

Bone marrow analysis should include an aspirate for cellular morphology, cytogenetic analysis and flow cytometry, and a core biopsy for bone marrow cellularity. If it is not possible to conduct cytogenetic analysis or flow cytometry on the bone marrow aspirate, then attempts should be made to carry out the tests on a blood sample. Full reports must be provided by the investigator for documentation on the Patient Safety database.

#### 6.4.12 Physical examination

For timing of individual measurement refer to study schedule (<u>Table 1</u>, <u>Table 2</u>, and <u>Table 3</u>). A physical examination will be performed according to site's local practice.

Clinical signs and symptoms of disease recurrence should be further investigated as appropriate (please refer to Section 6.3).

# 6.4.13 ECG

# 6.4.13.1 Resting 12-lead ECG

ECGs are required during screening within 28 days prior to randomisation.

Twelve-lead ECGs will be obtained after the patient has been rested in a supine position for at least 5 minutes. The investigator or designated physician will review the paper copies of each of the timed 12-lead ECGs.

NCI Version Date: 05-06-2021 110(177) NSABP B-55/BIG 6-13

ECGs will be recorded at 25 mm/sec. All ECGs should be assessed by the investigator as to whether they are clinically significantly abnormal / not clinically significantly abnormal. If there is a clinically significant abnormal finding, the investigator will record it as an AE on the eCRF. The original ECG traces must be stored in the patient medical record as source data.

# 6.4.14 Vital signs

Height will be assessed at screening only.

Weight will be assessed at screening and as clinically indicated at any other time.

Any changes in vital signs should be recorded as an AE, if applicable.

The date of collection and measurement will be recorded on the appropriate eCRF.

# 6.4.14.1 Pulse and blood pressure

Blood pressure and pulse rate will be measured preferably using a semi-automatic BP recording device with an appropriate cuff size. For timings of assessments refer to the Study Schedule (see Table 1 and Table 2).

The date of collection and measurement will be recorded on the appropriate eCRF.

# **6.4.14.2** Body temperature

Body temperature will be measured in degrees Celsius at the times indicated in the Study Schedule (see <u>Table 1</u> and <u>Table 2</u>).

The date of collection and measurement will be recorded on the appropriate eCRF.

# 6.4.15 Other safety assessments

# 6.4.15.1 Serum or urine pregnancy test

Pregnancy tests on serum or urine samples will be performed for women of childbearing potential within 28 days prior to randomisation (<u>Table 1</u>), on Day 1 of the study prior to commencing treatment, at the time points shown in <u>Table 2</u> during study treatment and at the 30 day follow up visit. Tests will be performed by the hospital's local laboratory. If results are positive the patient is ineligible/must be discontinued from study treatment immediately. Details of the pregnancy tests must be recorded in the patient's medical records.

# 6.5 Patient reported outcomes (PRO)

# 6.5.1 FACIT-Fatigue

The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F Scale) is a 13-item questionnaire that assesses patient self-reported fatigue and its impact upon daily activities and function (Yellen et al 1997). Response options for each item range from 0 (Not at all) to 4 (Very much), where higher scores indicate greater patient-reported fatigue. The FACIT-F scale was originally developed to evaluate fatigue associated with anaemia in cancer patients and has been used as an endpoint in clinical trials in various cancer populations including breast cancer

NCI Version Date: 05-06-2021 111(177) NSABP B-55/BIG 6-13
and non-small cell lung cancer. Content validity of the FACIT-F has been demonstrated in a large sample of mixed cancer patients (n>300). Reliability (internal consistency, test-retest reliability, criterion validity, and responsiveness/sensitivity to change) of the FACT-F has also been documented (Yellen et al 1997).

#### **6.5.2 EORTC QLQ-C30**

In this study patient-reported disease related symptoms and health-related quality of life (HRQoL) will be evaluated using the validated EORTC QLQ-C30 questionnaire (<u>Aaronson et al 1993</u>). The EORTC QLQ-C30 questionnaire was developed to assess HRQoL and is the most commonly used cancer-specific tool in oncology. It has undergone extensive testing and validation as well as detailed cross-cultural testing and validation and has been used in breast cancer trials.

The EORTC QLQ-C30 comprises 30 questions designed for all cancer types. Questions can be grouped into the following subscales:

- 5 multi-item functional scales (physical, role, emotional, cognitive and social functioning)
- A 2-item global health status scale
- Symptom scales/items
  - -3 multi-item symptom scales (fatigue, pain, nausea vomiting)
  - -Dyspnoea
  - -Insomnia
  - -Appetite loss
  - -Constipation
  - -Diarrhoea
  - Financial difficulties

#### 6.5.3 Administration of PRO questionnaires

FACIT-Fatigue and EORTC QLQ-C30 questionnaires will be collected at baseline (within screening period after eligibility confirmed but prior to randomisation) and then 6 months, (24 weeks), 12 months (52 weeks), 18 months and 24 months following randomisation.

Questionnaires shall be administered to a patient by delegated site personnel (e.g., a research nurse, study coordinator) adequately trained and listed on Site's Delegation Log. Site shall assign a trained back-up person to cover if that individual is absent. The significance and relevance of the data need to be explained carefully to participating patients so that they are motivated to comply with data collection.

The instructions for completion of the PRO questionnaires are as follows:

NCI Version Date: 05-06-2021 112(177) NSABP B-55/BIG 6-13

- They must be completed at the clinical visit prior to any other study procedures (following informed consent) and before discussion of disease progress to avoid biasing the patient's responses to the questions. They must be completed in private by the patient
- The patient should be given sufficient time to complete at their own speed
- The patient should not receive help from relatives, friends or clinic staff to answer the questionnaire. However, if the patient is unable to read the questionnaires (e.g., is blind or illiterate) the questionnaires may be read out by trained clinic staff and responses recorded
- On completion of the questionnaires they should be handed back to the person responsible for questionnaires who should check for completeness
- Only one answer should be recorded for each question.

Completed questionnaires must be faxed to the NRG Oncology SDMC (see <u>Information Resources</u>).

After the baseline, questionnaires are to be administered at follow-up visits, so that when a follow-up visit is delayed, completion of the questionnaire may also be delayed. Patients who experience disease recurrence or diagnosis of a second primary cancer will not be expected to continue with the PRO assessments. Patients who discontinue study drug for other reasons will be expected to continue the PRO assessments per protocol schedule if they have not indicated study withdrawal. Patients who never initiate study medication should not continue to complete PRO assessments. If a patient declines to complete a scheduled PRO assessment or if the questionnaire is not completed for any other reason (and cannot be completed by phone or mail), a Quality of Life Missing Data form should be submitted by the institution instead.

#### 6.5.4 Reimbursement

All sites will receive reimbursement for the PRO study from funding provided by AstraZeneca. Cancer Control credits will not be available.

#### 6.6 Biomarkers

Tumour and blood samples will be collected for mandated and optional biomarker work as detailed in the B-55/6-13 Pathology and Correlative Science Instructions.

For blood volume see Section 7.1

#### 6.6.1 Biomarker samples

The archival diagnostic tumour sample is mandated\* and the screening blood samples for *BRCA* mutation status are mandated.

NCI Version Date: 05-06-2021 113(177) NSABP B-55/BIG 6-13

 Table 12
 Samples for Biomarker Research

| Sample Type | Visits | Optional or Mandatory |
|---|---|---|
| Whole blood sample for prospective germline <i>BRCA</i> testing at central laboratory for patients with unknown <i>BRCA</i> status and for confirmation of <i>BRCA</i> status for those with previous results | Screening | Mandatory |
| Whole blood sample for assessment of current and future <i>BRCA</i> mutation assay(s) | Screening | Mandatory |
| Archival tumour sample Surgical tumour samples for adjuvant patients | Screening | Mandatory* for all randomised patients |
| Pre-treatment diagnostic core biopsy for neoadjuvant patients | Screening | Required* for all randomised patients |
| Surgical tumour sample post neoadjuvant chemotherapy | Screening | Required* for all randomised neoadjuvant patients |
| On-study disease recurrence tumour biopsy | At disease recurrence | Optional |
| Blood samples (plasma and serum) for biomarker analysis | Day 1 prior to first dose<br>of study treatment, 30<br>days post study treatment<br>discontinuation, disease<br>recurrence | Mandatory |
| Redacted | | |

\*For adjuvant patients, this refers to the surgical specimen; for neoadjuvant patients, both the pretreatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required.

The tumour and blood samples collected in this study will be used for studies specified in the B-55/6-13 protocol and for studies to be conducted in the future related to the purposes of the B-55/6-13 study and not currently described in the protocol document.

Detailed protocols for the genomics work described in this protocol will be developed as separate protocols to include analytical and statistical methodologies and will be submitted for review and approval of these methodologies in accordance with the National Clinical Trials Network. Studies conducted in the future related to the purposes of the B-55/6-13 study and not currently

NCI Version Date: 05-06-2021 114(177) NSABP B-55/BIG 6-13

described in the protocol document will be submitted for review and approval in accordance with the National Clinical Trials Network.

The samples and data from this research will be coded and not identified with any personal details. Each sample will be identified with the B-55/6-13 Patient ID number. In this way biomarker data may be correlated with clinical data, samples destroyed in the event of withdrawal of consent and regulatory audit enabled. However, only the investigator will be able to link the biomarker sample to the individual patient. Research biomarker data may be generated in real time during the study or retrospectively and will have unknown clinical significance. The study investigative team will not provide research biomarker results to patients, their family members, any insurance company, an employer, clinical study investigator, general physician or any other third party unless required to do so by law. The patient's samples will not be used for any purpose other than those described in the protocol.

The *gBRCA* status result from the Myriad assessment for patients with unknown *BRCA* status will be provided to the investigator and will be collected as part of the patient's demography and medical history details.

#### 6.6.2 Collection of blood sample for Myriad germline BRCA1 and BRCA2 testing

Two blood samples are mandated for all patients. One sample will be used to test for *BRCA* mutations using the current commercial Myriad BRCAnalysis test. This result will confirm or determine patient eligibility. The second sample is required for a bridging study to validate the companion diagnostic test for olaparib (see Section 6.6.2.1 below).

All patients must have a known deleterious or suspected deleterious germline *BRCA* mutation to be randomised; this may have been determined by local genetic testing prior to study entry or may be assessed as part of the enrolment procedure for the study (via a central testing by Myriad), see Section 6.2.1. The specific gBRCA alteration on which eligibility is based must be entered into the trial database by selecting the appropriate value from the drop down menu. If the central laboratory analysis does not confirm a local gBRCA determination, that information should also be entered in the eCRF, along with indication of whether or not the patient was enrolled into the trial.

Residual blood (or its derivatives) may be used to evaluate future BRCA companion diagnostic tests and for additional exploratory work, to elucidate the mechanism of response, understand the mode of action of study treatment, and improve the understanding of disease recurrence (including BRCA mutation status and its role in response).

For blood volume see Section 7.1.

# 6.6.2.1 Collection of a blood sample for assessment of current and future *BRCA* mutation assay(s)

At the time that the sample is collected for shipment to Myriad for central testing, all patients will be required to provide a second mandatory 9 ml blood sample that will be stored for subsequent assessment of current and future *BRCA* mutation assay(s).

NCI Version Date: 05-06-2021 115(177) NSABP B-55/BIG 6-13

Samples may also be used to investigate future *BRCA* mutation assays as well as mutations in other genes known/predicted to have a role in breast cancer.

Please refer to the B-55/6-13 Pathology and Correlative Science Instructions for further details of archival tumour collection, shipping and storage.

| Redacted | Redacted | |
|----------------------|----------|---|
| Redacted | | |
| Redacted | | |
| Redacted | | |
| Redacted | | |
| reducted | | |
| | | 7 |
| Redacted | Padastad | |
| Redacted | Redacted | |
| Redacted | Redacted | |
| Redacted<br>Redacted | Redacted | |
| Redacted<br>Redacted | Redacted | |
| Redacted<br>Redacted | Redacted | |
| Redacted | Redacted | |
| Redacted | Redacted | |
| Redacted | Redacted | |
| Redacted | Redacted | |
| Redacted | Redacted | |
| Redacted | Redacted | |





# 6.8 Pharmacokinetics (Optional)

PK sampling will not be done in the US.

PK sampling (optional) is to be performed in a subset of patients. Each patient participating in this component of the study will be asked to provide 5 blood samples, one from each of the pre-defined time windows below, preferably on visit 4, day 29. Nevertheless, the samples can also be taken at a later treatment visit, provided that PK consent was obtained beforehand.

- Pre-dose (before morning dose)
- Between 0 and 0.5 hours post-dose
- Between > 0.5 and 1.5 hours post-dose
- Between 3 and 6 hours post-dose
- Between > 6 and 12 hours post dose (before evening dose)

# 6.8.1 Pharmacokinetic samples (Subset of patients)

Approximately 150 patients randomised to olaparib/placebo, at pre-agreed sites will have PK assessment samples taken. PK sampling will not be done in the US.

#### 6.8.2 Collection of samples

PK samples are to be taken as a blood sample (2 mL) for determination of olaparib concentrations in plasma. It is essential that PK blood sampling is conducted within the protocol sample collection windows indicated above.

To ensure that the assessments are carried out in the correct order, and that PK sampling is conducted within the required sampling window, it will be necessary to arrange the assessment procedures so that the PK assessments fall on/around the correct timing (see <u>Section 6.8</u>). The actual time of dosing and collection of all PK samples must be recorded as described below:

It is essential that the time of all 5 PK samples is recorded and that the times of the morning and evening dose on the day of PK sampling and the time of dose the evening before is recorded.

For blood volume see Section 7.1.

NCI Version Date: 05-06-2021 118(177) NSABP B-55/BIG 6-13

#### 6.8.3 Determination of drug concentration

Samples for determination of olaparib concentrations in plasma will be analysed by Covance on behalf of Clinical Bioanalysis Alliance, AstraZeneca R&D, using an appropriate bioanalytical method. Full details of the analytical method used will be described in a separate bioanalytical report. Placebo samples will not be analyzed unless specified.

#### 6.9 Health economics

# 6.9.1 Resource use (serious adverse events)

Resource use for serious adverse events (including hospitalisations) will be captured through the adverse reporting procedures described in <u>Section</u> <u>6.4</u>.

#### 7. BIOLOGICAL SAMPLING PROCEDURES

#### 7.1 Volume of blood

The volume of blood that will be drawn from each patient will vary, dependent upon the length of time that the patient remains in the trial and if the patient is in the subset having PK samples taken. However, the total volume of blood to be drawn from each patient in the study (including for PK samples), assuming they complete screening, 12 months of treatment, a treatment discontinuation visit and the 30-day follow-up visit, should not exceed 208 mL.

Safety laboratory assessments will be performed locally at each centre's laboratory by means of their established methods. The number of samples/blood volumes is therefore subject to site-specific change.

Extra blood samples may also be collected if, for example, additional samples are required for repeat safety assessments or *BRCA* testing.

The total volume of blood that will be drawn from each patient in this study is as follows:

Table 13 Volume of blood to be drawn from each patient

| Assessment | | Sample volume (mL) | No. of samples | Total volume (mL) |
|---|---|---|---|---|
| Safety | Clinical chemistry | 5 | 13 | 65 |
| | Haematology | 5 | 13 | 65 |
| | Coagulation | 5 | 1 | 5 |
| Whole blood sample to (retrospective/prosp | for Myriad <i>BRCA</i> test etive) | 9 | 1 | 9 |
| Whole blood sample current and future <i>BR</i> | | 9 | 1 | 9 |
| Redacted | | • | • | |

NCI Version Date: 05-06-2021 119(177) NSABP B-55/BIG 6-13

| Assessment | Sample volume (mL) | No. of samples | Total volume (mL) |
|---|---|---|---|
| Redacted | | | |
| | • | | |
| | • | | |
| | • | | |
| | _ | _ | _ |
| | • | • | • |
| Redacted | | | |
| | • | | I |
| Pharmacokinetic (Blood samples processed to plasma & frozen) (Optional) | 2 | 5 | 10 |
| Total | | | 208 |

# 7.2 Handling, storage and destruction of biological samples

The samples may be used up, disposed of after analyses or retained for further use as described here.

Biological samples for future research will be retained at the study bio-repository for a maximum of 15 years following the Last Patient's Last Visit in the study. The results from future analysis will not be reported in the Clinical Study Report but separately in a Scientific Report.

Biosamples collected for this study will be stored in study specific bio-repositories that are under the guardianship of BIG (non-US samples) and NRG Oncology and NCI (US samples) on behalf of the study Steering Committee.

#### 7.2.1 Pharmacogenetic samples

The processes adopted for ensuring confidentiality of samples for genetic analysis are important. Samples will be stored for a maximum of 15 years, from the date of the Last Patient's Last Visit, after which they will be destroyed. DNA is a finite resource that may be used up during analyses. Samples will be stored and used until no further analyses are possible or the maximum storage time has been reached.

DNA will be extracted from the blood sample. The DNA sample will be assigned a unique number replacing the information on the sample tube. Thereafter, the DNA sample will be identifiable by the unique DNA number only. The DNA number is used to identify the sample

and corresponding data at the AstraZeneca genetics laboratories, or at the designated contract laboratory. No personal details identifying the individual will be available to any person (AstraZeneca employee or contract laboratory staff working with the DNA.)

The samples and data for genetic analysis in this study will be single coded. The link between the patient enrolment/randomisation code and the DNA number will be maintained and stored in a secure environment, with restricted access within the Clinical Genotyping Group Laboratory Information Management System (LIMS) at AstraZeneca. The link will be used to identify the relevant DNA samples for analysis, facilitate correlation of genotypic results with clinical data, allow regulatory audit and to trace samples for destruction in the case of withdrawal of consent when the patient has requested disposal/destruction of collected samples not yet analysed.

#### 7.2.2 Pharmacokinetic samples

Pharmacokinetic samples will be disposed of after the Bioanalytical Report finalisation or six months after issuance of the draft Bioanalytical Report (whichever is earlier), unless requested for future analyses. Additional analyses may be conducted on the anonymised, pooled pharmacokinetic samples to further evaluate and validate the analytical method. Any results from such analyses will be reported separately from the Clinical Study Report (CSR).

Sample reproducibility analysis, if any, will be performed alongside the bioanalysis of the test samples. The results from the evaluation will not be reported in the CSR but separately in a Bioanalytical Report. Anonymised samples will be retained for no longer than 12 months after the Bioanalytical Report is finalised.

# 7.3 Labeling and shipment of biohazard samples

The Principal Investigator should ensure that samples are labelled and shipped in accordance with the B-55/6-13 Pathology and Correlative Science Instructions and the Biological Substance, Category B Regulations (materials containing or suspected to contain infectious substances that do not meet Category A criteria), see <u>Appendix B</u> 'IATA 6.2 Guidance Document'.

Any samples identified as Infectious Category A materials should not be shipped and no further samples will be taken from the patient unless agreed with AstraZeneca/NRG Oncology/BIG or partners and appropriate labelling, shipment and containment provisions are approved.

# 7.4 Chain of custody of biological samples

A full chain of custody is maintained for all samples throughout their lifecycle.

The Principal Investigator at each centre is responsible for ensuring full traceability of collected biological samples from the patients while in storage at the centre until shipment or disposal (where appropriate).

The sample receiver keeps full traceability of the samples while in storage and during use until used or disposed of or until further shipment and keeps documentation of receipt of arrival.

NCI Version Date: 05-06-2021 121(177) NSABP B-55/BIG 6-13

AstraZeneca/NRG Oncology/BIG and their Partners keep oversight of the entire life cycle through internal procedures, monitoring of study sites and auditing of external laboratory providers.

Biosamples collected for this study will be stored in study specific bio-repositories that are under the guardianship of BIG (non-US samples) and NRG Oncology and NCI (US samples) on behalf of the study Steering Committee.

Samples retained for further use are registered in the bio-repositories systems during the entire sample life cycle.

If required, the remaining biological samples are returned to the site, according to local regulations or at the end of the retention period, whichever is the sooner.

#### 7.5 Withdrawal of informed consent for donated biological samples

If a patient withdraws consent to the use of donated biological samples, the samples will be disposed of/destroyed, and the action documented. If samples are already analysed, AstraZeneca/NRG Oncology/BIG and their Partners are not obliged to destroy the results of this research.

*BRCA* sample: As collection of the biological samples is an integral part of the study, then the patient is withdrawn from further study participation.

Archival tumour sample: Although mandatory\*, the patient may continue in the study if the patient is already randomised.

\*For adjuvant patients, this refers to the surgical specimen; for neoadjuvant patients, both the pre-treatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3 mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required.

Tumour samples at relapse: As collection of the biological samples is an optional part of the study, then the patient may continue in the study.

Pharmacokinetic samples: As collection of the pharmacokinetic samples is an optional part of the study, then the patient may continue in the study.

Blood samples for biomarker analysis (e.g. cfDNA): Collection of the biological samples is a mandatory part of the study, however, the patient may continue in the study despite withdrawing consent for analysis of the biomarker samples.

NCI Version Date: 05-06-2021 122(177) NSABP B-55/BIG 6-13

The Principal Investigator/site staff:

- Should ensure that NRG SDMC is notified immediately of a patients' withdrawal of informed consent for the use of donated samples
- Should ensure that biological samples from that patient, if stored at the study site, are immediately identified, disposed of /destroyed, and the action documented
- Should ensure that the laboratory(ies) holding the samples is/are informed about the withdrawn consent immediately and that samples are disposed/destroyed, the action documented and the signed document returned to the study site
- Should ensure that the patient and study representative are informed about the sample disposal.

The study representative ensures that the central laboratory(ies) holding the samples is/are informed about the withdrawn consent immediately and that samples are disposed of/destroyed and the action documented and returned to the study site.

# 8. ETHICAL AND REGULATORY REQUIREMENTS

# 8.1 Ethical conduct of the study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/Good Clinical Practice, applicable regulatory requirements and the AstraZeneca policy on Bioethics and Human Biological Samples.

#### 8.2 Patient data protection

The Informed Consent Form will incorporate (or, in some cases, be accompanied by a separate document incorporating) wording that complies with relevant data protection and privacy legislation.

AstraZeneca will not provide individual genotype results to patients, any insurance company, any employer, their family members, general physician or any other third party, unless required to do so by law.

Extra precautions are taken to preserve confidentiality and prevent genetic data being linked to the identity of the patient. In exceptional circumstances, however, certain individuals might see both the genetic data and the personal identifiers of a patient. For example, in the case of a medical emergency, a study medical representative or an investigator might know a patient's identity and also have access to his or her genetic data. Also Regulatory authorities may require access to the relevant files, though the patient's medical information and the genetic files would remain physically separate.

NCI Version Date: 05-06-2021 123(177) NSABP B-55/BIG 6-13

The exception to the above is the result of the Myriad gBRCA test. This will be made available to the Investigator and patient.

# 8.3 Ethics and regulatory review

An IRB must approve the final study protocol, including the final version of the Informed Consent Form and any other written information and/or materials to be provided to the patients. The investigator will ensure the distribution of these documents to the applicable IRB, and to the study site staff.

The opinion of the IRB should be given in writing. The investigator should submit the written approval to the CTSU before enrolment of any patient into the study.

The IRB should approve all advertising used to recruit patients for the study.

AstraZeneca/BIG/Partners (and NRG Oncology/CTEP for US centres) should approve major modifications to the Informed Consent Form that are needed to meet local requirements.

If required by local regulations, the protocol should be re-approved by the IRB annually.

Before enrolment of any patient into the study, the final study protocol, including the final version of the Informed Consent Form must be approved by a local IRB or the NCI Central Institutional Review Board (CIRB), according to local regulations.

NRG Oncology will handle the distribution of these documents to the national regulatory authorities.

AstraZeneca/BIG/Partners will provide Regulatory Authorities, IRBs/Ethics Committees and Principal Investigators with safety updates/reports according to local requirements, including SUSARs (Suspected Unexpected Serious Adverse Reactions), outside the United States, where relevant. NRG Oncology will determine distribution of safety updates/reports as appropriate, in the United States.

Each Principal Investigator is responsible for providing the IRB with reports of any serious and unexpected adverse drug reactions from any other study conducted with the investigational product according to local requirements. If applicable, AstraZeneca will provide this information to the Principal Investigator so that he/she can meet these reporting requirements.

#### 8.4 Informed consent

The Principal Investigator(s) at each centre will:

- Ensure each patient is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study
- Ensure each patient is notified that they are free to discontinue from the study at any time
- Ensure that each patient is given the opportunity to ask questions and allowed time to consider the information provided

NCI Version Date: 05-06-2021 124(177) NSABP B-55/BIG 6-13

- Ensure each patient provides signed and dated informed consent before conducting any procedure specifically for the study
- Ensure the original, signed Informed Consent Form(s) is/are stored in the Investigator's Study File
- Ensure a copy of the signed Informed Consent Form is given to the patient
- Ensure that any provisions for patients harmed as a consequence of study participation are described in the informed consent form that is approved by an IRB.

# 8.5 Changes to the protocol and informed consent form

Study procedures will not be changed without the mutual agreement of the International coordinating Investigator, National Co-ordinating Investigator, and the Principal Investigator and AstraZeneca/BIG/NRG Oncology/Partners and the study Steering Committee.

If there are any substantial changes to the study protocol, then these changes will be documented in a study protocol amendment and where required in a new version of the study protocol (Revised Clinical Study Protocol).

Any protocol amendment must be approved by the relevant IRB and if applicable, should obtain the national regulatory authority approval, before implementation. Local requirements are to be followed for amended protocols.

NRG Oncology will distribute any subsequent amendments and new versions of the protocol to each Principal Investigator(s). For distribution to IRBs see <u>Section</u> <u>8.3</u>.

If a protocol amendment requires a change to a centre's Informed Consent Form, AstraZeneca/BIG/Partners, NRG Oncology/CTEP for US centres, and the centre's IRB are to approve the revised Informed Consent Form before the revised form is used.

If required by local regulations, any administrative changes will be communicated to or approved by each IRB.

#### 8.6 Audits and inspections

Authorised representatives of NRG Oncology may perform audits or inspections at the centre, including source data verification. The purpose of an audit or inspection is to systematically and independently examine all study-related activities and documents, to determine whether these activities were conducted, and data were recorded, analysed, and accurately reported according to the protocol, Good Clinical Practice (GCP), guidelines of the International Conference on Harmonisation (ICH), and any applicable regulatory requirements. The investigator/site staff should contact the Protocol Officer immediately if contacted by a regulatory agency about an inspection at the centre.

NCI Version Date: 05-06-2021 125(177) NSABP B-55/BIG 6-13

#### 9. STUDY MANAGEMENT

# 9.1 Pre-study activities

Qualification visits are not performed by NRG Oncology. NRG Oncology Member Institutions must determine that the sites are appropriate for the study. NRG Oncology distributes the approved protocol to its member institutions which are in good standing. Those sites which are confident that they have significant investigator interest and available patients proceed by seeking local (or central) Institutional Review Board approval. Upon receipt of the approval, a database of site IRB approvals is maintained through the NCI CTSU. Patient entry cannot proceed unless an up-to-date IRB approval is in this database.

# 9.2 Training of study site personnel

The Principal Investigator should ensure that appropriate training relevant to the study is given to all site staff, and that any new information relevant to the performance of this study is forwarded to the staff involved.

The Principal Investigator will maintain a record of all individuals involved in the study (medical, nursing and other staff).

# 9.3 Monitoring of the study

The study will be monitored by site audit visits, submission of copies of source documents for centralized review, and communication with the investigator and appropriate staff by NRG Oncology to:

- Provide information and support to the investigator(s)
- Confirm that facilities remain acceptable
- Confirm that the investigational team is adhering to the protocol, that data are being accurately and timely recorded in the eCRFs, that biological samples are handled in accordance with the B-55/6-13 Pathology and Correlative Science Instructions and that study drug accountability checks are being performed
- Perform source data verification (a comparison of the data in the eCRFs with the patient's medical records at the hospital or practice, and other records relevant to the study) including verification that the appropriate version of the consent form was used and that it was signed and dated prior to any study procedures. This will require direct access to all original records for each patient (e.g. clinic charts)
- If relevant, ensure withdrawal of informed consent to the use of the patient's biological samples is reported and biological samples are identified and disposed of/destroyed accordingly, and the action is documented, and reported to the patient.

NCI Version Date: 05-06-2021 126(177) NSABP B-55/BIG 6-13

The investigator will provide direct access to source data/documents for audits, IRB review, and regulatory inspections. NRG Oncology will be available between visits if the investigator(s) or other staff at the centre needs information and advice about the study conduct.

# 9.4 Study timetable and end of study

The end of the study is defined as 'the last visit of the last patient undergoing the study'.

The study is expected to start in Q1 2014 and to end by 2028.

The study will end approximately 10 years following the randomisation of the last patient. Patients will be followed up until 10 years after the randomisation of the last patient.

The study may be prematurely terminated at individual centres if the study procedures are not being performed according to GCP, or if recruitment is slow. AstraZeneca may also terminate the entire study prematurely upon recommendations of the study IDMC if concerns for safety arise within this study or in any other study with olaparib.

#### 10. DATA MANAGEMENT

Data management will be performed by the NRG Oncology SDMC.

The data collected through third party sources will be obtained and reconciled against study data by Frontier Science.

Adverse events and medical/surgical history will be classified according to the terminology of the latest version of the Medical Dictionary for Regulatory Activities (MedDRA). Medications will be classified according to the AstraZeneca Drug Dictionary. Coding will be done by Frontier Science.

Additional details of data management procedures can be found in the Data Management Plan for the Study. This document will be continuously updated through the life of the study.

Data queries will be raised for inconsistent, impossible or missing data. All entries to the study database will be available in an audit trail.

The data will be validated as defined in the Data Management Plan. Quality control procedures will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. The Data Management Plan will also document the roles and responsibilities of the various functions and personnel involved in the data management process.

When all data have been coded, validated, and locked, clean file will be declared. Any treatment revealing data may thereafter be added and the final database will be locked.

The results from genetic research may be reported in the CSR for the main study, or in a separate report as appropriate. Refer to  $\underline{\text{Appendix } C}$ .

NCI Version Date: 05-06-2021 127(177) NSABP B-55/BIG 6-13

#### 11. EVALUATION AND CALCULATION OF VARIABLES

# 11.1 Calculation or derivation of efficacy variable(s)

#### 11.1.1 Primary endpoint

The primary endpoint of the trial is invasive disease free survival (IDFS), defined as the time from randomisation to date of first recurrence, where recurrence is defined as loco-regional, distant recurrence, new cancer or death from any cause. IDFS is further detailed according to the standardised STEEP system definition (Hudis et al 2007) as one of the following:

- Ipsilateral invasive breast tumour recurrence (IIBTR): Invasive breast cancer involving the same breast parenchyma as the original primary.
- Regional invasive breast cancer recurrence: Invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast.
- Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or radiologically diagnosed as recurrent invasive breast cancer.
- Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
- Contralateral invasive breast cancer.
- Second primary non-breast invasive malignancies (i.e., excluding new in situ carcinomas
  of any site). Second primary non-breast invasive malignancies include hematologic
  malignancies and MDS. Squamous or basal cell skin cancers will not be counted as
  primary endpoint events.

Loco-regional recurrence of the disease (ipsilateral or regional invasive breast cancer) should be cytologically/histologically confirmed. Appropriate imaging (CT, MRI bone and/or PET scan) of the chest/abdomen/pelvis or any other area as clinically indicated should be performed at the time of local recurrence to exclude further spread of the disease. Distant recurrence should be diagnosed by radiological examination and/or histopathological confirmation when metastatic lesion is easily accessible for biopsy.

For confirmed local recurrence events, the earliest date of diagnosis based on an objective finding (physical exam, radiological/imaging assessment, cytological/histopathological assessment) will be used to determine the time to event for the analysis but not the date of the first symptoms or blood analysis abnormality. For example if a physical exam results in 'suspected' disease recurrence and disease recurrence is then confirmed by cytology/histology then the date of the physical exam will be used to derive the time to event.

For confirmed distant recurrence the date of the earliest radiological/imaging examination or cytological/histopathological assessment linked to the diagnosis will be used to determine the

NCI Version Date: 05-06-2021 128(177) NSABP B-55/BIG 6-13

time to event for the analysis (i.e. physical exam will not be considered within the derivation of time to distant recurrence nor will be symptoms or blood analysis).

Invasive contralateral breast cancer or invasive non-breast secondary primary cancer should be confirmed by histopathological report. The date of the earliest objective finding related to diagnosis of the new cancer will be used as the date of new cancer for the analysis.

If two recurrence events (local and distant) are reported within 2 months of each other then this is referred to as a simultaneous event and will be considered as a single event. In this situation the worst case will be taken as the event 'type' but the date of recurrence will be the earliest date of the two events. For example if local and distant recurrence are reported within a 2 month period then for the analysis and reporting of IDFS the event type will be distant recurrence but the date of recurrence will be the earliest date of the two events.

If two recurrence events are reported but more than 2 months has elapsed between the events then the events will be regarded as two separate recurrence events and the earliest event and corresponding date of event will be used in the derivation of IDFS (i.e. IDFS is based on the first recurrence event).

If a patient dies during the study with no documented disease recurrence or invasive contralateral breast cancer or invasive non-breast secondary primary cancer then death will be regarded as an event and the date of death will be used to determine the patients IDFS time.

Patients who have not had a recorded IDFS event at the time of the analysis will be censored at the date of their last disease evaluation. Disease evaluation includes mammogram and/or breast MRI (MRI preferred for patients younger than 50 years), other radiological/imaging examination or clinical examination (e.g. physical exam).

#### 11.1.2 Secondary endpoints

#### 11.1.2.1 Overall Survival

Overall survival is defined as the time from the date of randomisation until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.

#### 11.1.2.2 Distant disease free survival (DDFS)

DDFS will be defined as the time from randomisation until documented evidence of first distant recurrence of breast cancer. Distant recurrence will include the following events:

- Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or radiologically diagnosed as recurrent invasive breast cancer.
- Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
- Second primary non-breast invasive cancer.

NCI Version Date: 05-06-2021 129(177) NSABP B-55/BIG 6-13

Evidence of distant recurrence should be provided by either radiological examination or preferably by histopathological examination when metastasis is easily accessible for biopsy.

Second primary non-breast invasive cancer should be confirmed by histopathological report.

For the analysis of DDFS, the date of the confirmed DDFS event will use the earliest assessment date from the radiological and/or histological or cytological assessment. For example if a patient has distant recurrence suspected by radiological examination which is later confirmed by biopsy then the date of the radiological examination will be used as the date of event.

Patients who do not have documented evidence of DDFS at the time of the analysis of DDFS will be censored at the date of their last clinical examination (i.e. last physical exam or radiological evaluation).

The first site of distant recurrence will be recorded and used in the analysis. Information on subsequent sites of recurrence will also be collected during follow-up assessments to ensure as complete as possible information on distant recurrence is obtained.

# 11.1.2.3 Incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer

The incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer will each be considered separately and be defined as the number and percentage of patients with documented evidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer regardless of when this occurs (i.e. does not need to be their first recurrence event).

All patients should be followed for evidence of new primary breast cancers and all other cancers. This includes patients with a first event of local or distant recurrence as they may go on to develop new cancers in the future. All new cancers will be collected for all patients not just the first new cancer.

Data analyses of new contralateral breast cancer (invasive and non-invasive) will exclude patients who have had bilateral mastectomy prior to randomisation.

Data analyses of new ovarian cancers will exclude patients who have had both ovaries removed prior to randomisation.

Data analyses of new fallopian tube cancers will exclude patients who have had both fallopian tubes removed prior to randomisation.

Data analyses of new peritoneal cancer will include all patients in the ITT populations.

NCI Version Date: 05-06-2021 130(177) NSABP B-55/BIG 6-13

#### 11.2 Calculation or derivation of safety variable(s)

Safety and tolerability will be assessed in terms of AEs, deaths, laboratory data and vital signs. These will be collected for all patients. Appropriate summaries of these data will be presented as described in <u>Section 12</u>.

# 11.2.1 Other significant adverse events (OAE)

During the evaluation of the AE data, an AstraZeneca medically qualified expert will review the list of AEs that were not reported as SAEs and DAEs. Based on the expert's judgement, significant adverse events of particular clinical importance may, after consultation with the Global Patient Safety Physician, be considered OAEs and reported as such in the Clinical Study Report. A similar review of laboratory/vital signs/ECG data will be performed for identification of OAEs.

Examples of these are marked haematological and other laboratory abnormalities, and certain events that lead to intervention (other than those already classified as serious), dose reduction or significant additional treatment.

#### 11.3 Calculation or derivation of patient reported outcome variables

Patient reported outcomes will be assessed based on the FACIT-Fatigue symptoms and the EORTC QLQ-C30 questionnaires. Further details are given in <u>Section 12.2.3</u> and full details will be provided in the statistical analysis plan.

## 11.4 Calculation or derivation of pharmacokinetic variables

The pharmacokinetic (PK) analysis of the plasma concentration data for olaparib will be performed at AstraZeneca R&D or by a CRO identified by AstraZeneca R&D. The actual sampling times will be used in the PK calculations. For each patient providing a complete set of PK samples, non-linear mixed effects modelling (NONMEM) will be used to estimate steady state  $C_{max}$ , AUC and  $C_{min}$ .

#### 11.5 Calculation or derivation of pharmacodynamic variable(s) - not applicable

# 11.6 Calculation or derivation of Redacted variables

Any data summaries that will be reported in the main clinical study report will be detailed within the statistical analysis plan. Additional exploratory analyses or data summaries that may be produced outside of the main study report will be defined in an exploratory analysis plan, if appropriate.

#### 11.7 Calculation or derivation of health economic variables –not applicable

#### 12. STATISTICAL METHODS AND SAMPLE SIZE DETERMINATION

# 12.1 Description of analysis sets

A comprehensive statistical analysis plan (SAP) will be prepared before first subject in (FSI).

Table 14 gives a summary of outcome variables and analysis populations.

NCI Version Date: 05-06-2021 131(177) NSABP B-55/BIG 6-13

#### 12.1.1 Full analysis set

Intention to treat (ITT): The primary statistical analysis of the efficacy of olaparib will include all randomised patients and will compare the treatment groups on the basis of randomised treatment, regardless of the treatment actually received. Patients who were randomised but did not subsequently go on to receive study treatment are included in the Full Analysis Set (FAS).

For the interim analysis two efficacy populations will be defined.

- 1. ITT population: This will include all randomised patients and will compare the treatment groups on the basis of randomised treatment, regardless of the treatment actually received. Note: it is anticipated that all patients will be randomised by the time of the interim analysis.
- 2. Mature cohort ITT population: This will include the first 900 randomised patients only and will compare the treatment groups on the basis of randomised treatment, regardless of the treatment actually received.

#### 12.1.2 Safety analysis set

All patients who received at least one dose of randomised study treatment, olaparib or placebo, will be included in the safety analysis set. If a patient receives at least one dose of olaparib he/she will be summarised in the olaparib arm for safety summaries (e.g. olaparib arm will include patients randomised to olaparib who receive at least one dose of olaparib or placebo patients who receive at least one dose of olaparib in error at any time). If a patient randomised to olaparib receives only placebo treatment then he/she will be summarised as part of the placebo arm.

Table 14 Summary of Outcome Variables and Analysis Populations

| Outcome Variable | Populations |
|---|---|
| Efficacy Data - Interim | |
| IDFS | FAS (ITT), Mature cohort ITT |
| Other efficacy variables | FAS (ITT) |
| Efficacy data- Final | FAS (ITT) |
| IDFS, OS, DDFS, incidence of contralateral breast cancers, new primary ovarian, new primary fallopian tube cancers and new primary peritoneal cancer and symptom/HRQoL endpoints | |
| Demography | FAS (ITT) |
| Pharmacokinetics data | PK |
| Safety Data | |
| Exposure | Safety |
| Adverse Events | Safety |
| Lab measurements | Safety |
| Vital Signs | Safety |

NCI Version Date: 05-06-2021 132(177) NSABP B-55/BIG 6-13

#### 12.1.3 PK Analysis set

PK data will be analysed according to treatment received. This population will comprise all randomised to olaparib patients who receive at least one dose of study treatment and have at least one PK sample collected.

#### 12.2 Methods of statistical analysis

#### 12.2.1 Analysis of primary endpoint

#### 12.2.1.1 Primary analysis

The primary analysis of IDFS will occur when a minimum of 330 IDFS events have been observed (to provide at least 90% power to detect a hazard ratio of 0.7). Based on the event rate from the 10 November 2017 database, the number of IDFS events required to trigger the primary analysis is expected to be accrued by November 2020 (80% CI: March 2020 to September 2021). The maturity rate will be 18.3%, where maturity is defined as the number of events divided by the total number of randomised patients.

IDFS will be compared across two treatment arms using a log rank test stratified by the stratification factors at randomisation, and the corresponding p-value will be reported as the primary analysis result. In addition, IDFS will be analysed using a stratified Cox proportional hazard model stratified by the stratification factors at randomisation and using the Efron approach for handling ties. The point estimate of the treatment effect, i.e., the hazard ratio of IDFS (olaparib vs. placebo) will be obtained by maximizing the Cox partial likelihood function, which is the product of the partial likelihood of each stratum. The 95% confidence interval will be estimated using the profile likelihood approach.

A Kaplan-Meier plot of IDFS will be presented by treatment group. Summaries of the number and percentage of patients experiencing an IDFS event, and the type of event (recurrence or death) will be provided for each treatment.

The estimated 3 year IDFS will be summarised (using estimates from the KM curve) and presented by treatment group.

# 12.2.1.2 Sensitivity analysis

If applicable, an analysis will be performed for IDFS using the same model as described above but based on all randomised patients confirmed to have *gBRCA* mutations by the central test. This analysis is only required if the analysis population differs from the primary ITT population.

Any patients mis-stratified in the randomisation system (i.e. incorrect details are entered at the time of randomisation) will be included in the primary stratified log rank test and Cox proportional hazard model using the baseline data collected from the randomisation system (Registration and Randomisation System). If > 5% of randomised patients are incorrectly stratified (i.e., randomisation system data does not match baseline data), then a sensitivity analysis will be performed for IDFS based on the (correct) baseline data collected in the eCRF. If the results of ER and PgR status from the local and central labs differ in >5% of randomised

NCI Version Date: 05-06-2021 133(177) NSABP B-55/BIG 6-13

patients, a sensitivity analyses will also be performed based on ER and/or PgR positive/HER2 negative and TNBC subsets as defined by the central laboratory testing.

The assumption of proportionality will be assessed. Proportionality will be tested firstly by producing plots of complementary log-log (event times) versus log (time) and, if these raise concerns, a time dependent covariate would be fitted to assess the extent to which this represents random variation. Note that in the presence of non-proportionality, the HR will be interpreted as an average HR over the observed extent of follow-up.

As patients will be randomised, imbalances in demographic factors between the treatment groups are not anticipated. However if any imbalances should occur, these additional demographic variables may be fitted into the stratified Cox model. The HR and associated confidence interval would be presented.

#### 12.2.1.3 Subgroup analysis

Subgroup analyses will be conducted to assess consistency of treatment effect across potential or expected prognostic factors, including the baseline stratification factors.

If there are too few results available for a meaningful analysis of a particular subgroup (it is not considered appropriate to present analyses where there are less than 5 events in either treatment group), the relationship between that subgroup and IDFS will not be formally analysed. In this case, only descriptive summaries will be provided.

The following subgroups are of primary interest:

- Hormone receptor status (ER and/or PgR positive and HER2 negative; TNBC)
- Neoadjuvant chemotherapy; adjuvant chemotherapy
- Prior platinum therapy for current breast cancer (Yes; No)
- BRCA mutation type (BRCA1; BRCA2; BRCA1/2 both)
- Hormone receptor status by prior chemotherapy setting (if there are sufficient events to split into the four groups)
  - ER and/or PgR positive with neoadjuvant chemotherapy
  - ER and/or PgR positive with adjuvant chemotherapy
  - ER and PgR negative with neoadjuvant chemotherapy
  - ER and PgR negative with adjuvant chemotherapy
- BRCA status by prior platinum therapy setting
  - BRCA1 with prior platinum therapy for current breast cancer

NCI Version Date: 05-06-2021 134(177) NSABP B-55/BIG 6-13

- BRCA1 with no prior platinum therapy for current breast cancer
- BRCA2 with prior platinum therapy for current breast cancer
- BRCA2 with no prior platinum therapy for current breast cancer

The following additional subgroups will also be analysed to assess consistency in treatment effect across a broader set of baseline characteristics known before start of study medication:

- Type of prior Neo/Adjuvant chemotherapy (anthracycline; taxane; anthracycline plus taxane)
- Type of breast surgery prior to randomisation (breast conservation; unilateral mastectomy; bilateral mastectomy)
- Bilateral Oophorectomy (Yes; No)
- Axillary nodal status at surgery prior to randomisation (Positive or negative for the post adjuvant patients only)
- CPS+EG score baseline (2, 3 or 4; 5 or 6 for the post neoadjuvant group only)
- Age at randomisation (< 50; 50-64;  $\ge 65$ )
- Race
- Sponsor (AZ; NRG Oncology)

Other baseline variables may also be assessed if there is clinical justification. These would be pre-defined within the SAP.

For each subgroup, the HRs (olaparib: placebo) and associated CIs will be calculated from a Cox proportional hazards model (using the Efron approach for handling ties) that contains the treatment term, factor and treatment-by-factor interaction term. The treatment effect HRs for each treatment comparison along with their confidence intervals will be obtained for each level of the subgroup from this single model. The HRs and 95% CIs will be presented on a forest plot including the HR and 95% CI from the overall population (using the primary analysis).

No adjustment to the significance level for testing subgroups will be made since all these subgroup analyses will be considered exploratory. The results would be used as supportive data for the primary analysis of IDFS based on all randomised patients.

#### 12.2.1.4 Analysis of interaction

The presence of quantitative interactions will be assessed by means of an overall global interaction test. This will be performed in the overall population by comparing the fit of a Cox proportional hazards model including treatment, all covariates (including stratification factors), and all covariate-by-treatment interaction terms, with one that excludes the interaction terms and will be assessed at the 2-sided 10% significance level. If a covariate does not have more than 20

NCI Version Date: 05-06-2021 135(177) NSABP B-55/BIG 6-13

events per level (of the covariate) it will be included as a covariate in the model, but the covariate-by-treatment interaction term will be omitted. If the fit of the model is not significantly improved then it will be concluded that overall the treatment effect is consistent across the subgroups.

If the global interaction test is found to be statistically significant, an attempt to determine the cause and type of interaction will be made. Stepwise backwards selection will be performed on the saturated model, whereby (using a 10% level throughout) the least significant interaction terms are removed one-by-one and any newly significant interactions re-included until a final model is reached where all included interactions are significant and all excluded interactions are non-significant. Throughout this process all main effects will be included in the model regardless of whether the corresponding interaction term is still present. This approach will identify the factors that independently alter the treatment effect and prevent identification of multiple correlated interactions.

Any quantitative interactions identified using this procedure will then be tested to rule out any qualitative interaction using the approach of <u>Gail and Simon 1985</u>.

#### 12.2.2 Analysis of secondary endpoints

#### OS and DDFS

OS and DDFS will be analysed at the time of the IDFS analysis as per the multiple testing procedure (MTP) outlined in <u>Section 12.2.5</u> and will use the same methodology and model as described above for the primary analysis of IDFS.

If applicable, a sensitivity analysis will be performed for DDFS and OS using the same model as described above for IDFS but based on all randomised patients confirmed to have *gBRCA* mutations by the central test. This analysis is only required if the analysis population differs from the primary ITT population Subgroup analyses will also be conducted for DDFS and OS based on the same subgroups described above for IDFS.

DDFS and OS will be analysed at the time of the primary analysis for IDFS (when 330 IDFS events are reported).

The final OS analysis will be conducted once the trial follow up is complete (i.e. 10 years from when the last patient is randomised, estimated 14 years from first patient randomised assuming recruitment of 5 years).

In addition another analysis will be performed half way between the primary IDFS analysis and the final overall survival analysis (estimated around 10 years from first patient randomised but timings will be driven by the primary IDFS analysis once known). At this time point both DDFS and OS will be analysed and some alpha will be reserved for formal hypothesis testing. IDFS may also be updated if more information is available but this would be considered a supportive update of the primary analysis and no alpha will be reserved for IDFS.

For details on alpha spend and how this will be allocated across the planned analyses see <u>Section</u> 12.2.6.

NCI Version Date: 05-06-2021 136(177) NSABP B-55/BIG 6-13

# Incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer

The actual number and percentage of patients with new contralateral breast cancers (invasive and non-invasive), new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancers will be presented. In addition a table summarising all reported new cancers (i.e. not just breast, ovarian, fallopian tube or peritoneal cancers) will also be produced.

As described in <u>Section 11.1.2.3</u>, patients who have had a bilateral mastectomy prior to randomisation will be excluded from the analysis of new contralateral breast cancers (invasive and non-invasive) and patients who have had a bilateral oophorectomy prior to randomisation will be excluded from the analysis of new ovarian cancers and patients who have had their fallopian tubes removed prior to randomisation will be excluded from the analysis of new fallopian tube cancers.

The cumulative incidence of new primary contralateral invasive breast, new primary contralateral non-invasive breast, new primary ovarian cancers, new primary fallopian tube cancers and new primary peritoneal cancers will be compared between treatment groups using competing risk analysis (Gray test, Fine and Gray 1999). Death will be considered a competing risk for each endpoint. In addition, bilateral mastectomy after randomization will be a competing risk for the contralateral breast cancer analyses, bilateral oophorectomy will be a competing risk for the new primary ovarian cancers analysis and removal of the fallopian tubes will be a competing risk for the new primary fallopian tube cancer analysis. Hazard ratios and 95% confidence intervals from competing risks regression analyses (Fine and Gray 1999) adjusted for treatment and the stratification factors will also be presented – more details of these analyses are given in the SAP (Edition 2).

#### Safety

Safety data will be summarised descriptively in terms of AEs, vital signs, clinical chemistry & haematology and physical exam and will include data from the treatment and safety follow-up period. Cumulative incidence plots may also be presented for specific adverse events or groups events of interest. Further information on the summary of safety data will be provided in the SAP.

#### 12.2.3 Analysis of patient reported outcomes

#### 12.2.3.1 Hypotheses and objectives

The hypotheses and measurement strategy focus on the fact that patients in the trial will be starting with significant decrements in HRQoL and high rates of symptoms at study entry (baseline) due to previous chemotherapy and local treatments (surgery with or without radiation therapy). All analyses of Patient Reported Outcomes will be conducted on ITT population as listed in <u>Table 14</u>. Therefore, the following hypotheses are proposed, based on the expected toxicities of olaparib.

NCI Version Date: 05-06-2021 137(177) NSABP B-55/BIG 6-13

#### **Primary hypothesis**

Patients receiving olaparib may experience greater fatigue severity during treatment than those receiving placebo as measured by the FACIT-Fatigue scale at 6 and 12 months after randomisation.

# **Secondary hypotheses**

- Patients receiving olaparib may experience greater GI symptoms (nausea, vomiting and diarrhea) severity during treatment than those receiving placebo as measured at 6 and 12 months after randomisation but no difference expected by 24 months after randomisation.
- There will be no difference in fatigue post discontinuation of study treatment as measured at 18 and 24 months.
- There will be no difference in QOL between the two treatment arms as measured by the global QOL score and other sub scales from the EORTC QLQ-C30 at 6, 12, 18 and 24 months after randomisation and patients will demonstrate improvements in functioning over time

# **Primary PRO objective**

To determine the effect of olaparib on patient-reported fatigue at 6 and 12 months after randomisation as measured by the FACIT-Fatigue symptoms questionnaire.

#### **Secondary PRO objectives**

- To determine the effect of olaparib on patient-reported GI symptoms (nausea, vomiting and diarrhea) over time at 6, 12, 18 and 24 months as measured by the EORTC QLQ-C30 scale.
- To determine the effect of olaparib on patient reported fatigue over time at 6, 12, 18 and 24 months as measured by the FACIT-Fatigue questionnaire.
- To determine if there will be a difference in QOL between the two treatment groups over time as measured by the 2 item global QOL score of the EORTC QLQ-C30 scale at 6, 12, 18 and 24 months and assess if patients demonstrate improvement in scores over time.
- To examine and compare the effect of olaparib over time on different functional sub scale scores as measured by the EORTC QLQ-C30 and assess if patients demonstrate improvement in functioning over time, with particular interest in the physical and emotional sub scales.

NCI Version Date: 05-06-2021 138(177) NSABP B-55/BIG 6-13

#### 12.2.3.2 Statistical considerations for patient reported outcomes

#### Statistical analyses

# Primary endpoint - Fatigue

For the primary hypothesis, the composite fatigue score (FACIT-Fatigue questionnaire) measured at 6 and 12 months after randomisation will be compared between the two treatment arms using analysis of covariance (ANCOVA) with adjustment for the corresponding baseline measurement. Separate analyses will be done for patients who have received prior neoadjuvant chemotherapy and patients who have received standard post-surgical adjuvant chemotherapy. Separate analyses are preferable because the timing of chemotherapy is expected to impact the fatigue outcome directly. Each comparison will be performed at the significance level of 0.05. No multiple comparisons adjustment will be employed since these outcomes evaluate the toxicity of the study treatment.

To further assess the effect of olaparib on fatigue over time (study treatment period and the year following) the composite fatigue score (FACIT-Fatigue questionnaire) measured at 6, 12, 18 and 24 months after randomisation will be compared between the two treatment arms using a mixed model for repeated measures (MMRM) analysis of all of the post baseline scores. The model will include treatment, time and treatment by time interaction as explanatory variables and baseline score and baseline by time interaction as covariates. The treatment by visit interaction will remain in the model regardless of significance. The adjusted mean change from baseline estimates for each treatment arm, difference in the adjusted mean change from baseline estimates between the arms and corresponding confidence intervals will be presented by time point. Plots of the adjusted means changes over time will also be presented.

#### **Secondary PRO endpoints**

A secondary analysis based on GI symptoms (nausea, vomiting and diarrhea) over time from the EORTC QLQ-C30 scale will be performed using the same MMRM model described above. The adjusted mean change from baseline estimates for each treatment arm, difference in the adjusted mean change from baseline estimates between the arms and corresponding confidence intervals will be presented by visit. Plots of the adjusted means changes over time will also be presented for nausea, vomiting and diarrhea.

To assess if there are any difference in HRQoL, the 2 item global QOL score assessed by EORTC QLQ-30 measured at 6, 12, 18 and 24 months after randomisation will be compared between the two treatment arms using the same MMRM model described above. Plots over time will also be produced for the global QOL score.

In addition, other subscales of the EORTC QLQ-C30 will be analysed using the MMRM model described above with particular interest in the emotional and physical subscales. Plots over time will also be produced.

All secondary analyses are considered exploratory and therefore no adjustments for multiplicity will be made. For each comparison, p-values (along with CIs) will be generated to help aid interpretation of the results using a nominal significance level of 0.05 (2-sided).

NCI Version Date: 05-06-2021 139(177) NSABP B-55/BIG 6-13

Because this trial is being conducted internationally, responses to patient reported outcomes may be influenced by differences between country/language categories (<u>Bernhard J et al 2007</u>). Therefore, analyses will be stratified by country/language groups. Further details will be provided in the SAP.

Adjustment for previous treatment exposures (radiation, type of chemotherapy, and surgery) may also be considered as part of the secondary analyses. Further details will be given in the SAP.

# Sample size consideration

We assume that half of triple negative patients and a quarter of hormone receptor positive patients will have received neoadjuvant chemotherapy and we anticipate that 95% of patients enrolled in the trial will complete the HRQoL instrument. In addition, adjusting downward to allow for 20% of missing data at the 12 months assessment point, we expect that data from 633 neoadjuvant and 735 adjuvant patients will be available (assuming that 15% of the total 1800 enrolled patients are ER and/or PgR positive HER2 negative). These will be sufficient to provide statistical power of 93% and 96% correspondingly to detect a difference of 3 points on the FACIT-Fatigue scale score between treatment groups assuming a standard deviation of 10.9 (Cella D et al 2002) (estimated SD of mean baseline score) and controlling  $\alpha$ -level at 0.05. The 3-point difference is the clinically meaningful difference reported by the developers of the scale (Cella D et al 2002), and we are hypothesizing that the olaparib arm will be worse. A collection of PROs and QOL from all patients enrolled in the main trial will give us sufficient statistical power to detect important differences between two treatment groups.

# **Missing PRO data**

A certain amount of missing data is expected. If data for individual items are missing, imputation will be done as follows: if less than 50% of the subscale items were missing (e.g. at most 2 out of 5 items, etc), the subscale score based on the non-missing items will be divided by the number of non-missing items and multiplied by the total number of items on the subscale. If at least 50% of the items are missing, that subscale will be treated as missing (not evaluable). If the scale is a single-item measure, a missing value will automatically be defined as 'Non-Evaluable'. The information from patients with missing data will be reviewed in order to determine whether data analytic procedures are likely to be biased. Patients with missing data will be reviewed for imbalances in factors such as trial arm, treatment adherence, institution, and reason for non-adherence. When QOL data are missing at a particular time point, data from prior time points will be reviewed in order to investigate whether missing status was preceded by a significant change in QOL scores. In addition, we will investigate whether missing item status is related to other scores on the same questionnaire. If no missing data mechanism can be detected following this review, the data will be analysed assuming the data are missing at random. If, on the other hand, a missing data mechanism appears to be present, we will undertake to develop an appropriate analytic strategy to control for the potential bias and, if possible, to impute the missing values. We will also present sensitivity analyses based on varying assumptions about the missing-data mechanism.

Full details on the analysis and derivation of PRO endpoints will be provided in the statistical analysis plan (SAP).

NCI Version Date: 05-06-2021 140(177) NSABP B-55/BIG 6-13

# 12.2.3.3 Pharmacokinetic analysis

The plasma concentration-time data will be analysed by non-linear mixed effects modelling in order to evaluate the pharmacokinetic characteristics of olaparib, quantify variability in the pharmacokinetics, identify demographic or pathophysiological covariates which may explain the observed variability and explore exposure-response relationships.

The olaparib plasma concentration data obtained from the samples collected in this study will be included in the listings of the CSR but these data will be pooled with data from other studies in order to perform a population PK analysis. The results of this analysis will be reported in a separate population PK report.

| Redacted | Redacted |
|----------|----------|
| Redacted | |
| Redacted | |

#### 12.2.5 Multiplicity strategy for primary and key secondary endpoints

The primary endpoint of the study is IDFS. However, key secondary endpoints will be OS and DDFS.

In order to describe the nature of the benefits of olaparib treatment IDFS, DDFS and OS will be tested at a 2-sided significance level of 5%.

However, in addition, in order to strongly control the overall type I error at 2.5% 1-sided, a multiple testing procedure (MTP) will be employed across the primary endpoint and all key secondary endpoints intended for label claims (DDFS and OS). The MTP will account for any interim analyses on IDFS, DDFS and OS and also planned further analyses post the primary IDFS analysis data cut off.

A hierarchical testing strategy will be employed where IDFS is tested first using the full test mass (i.e. full 2.5%, 1-sided alpha), then DDFS and OS will be tested if IDFS is significant based on a weighted proportion of the test mass (2% for DDFS and 0.5% for OS, 1-sided) which can be recycled to secondary endpoints not yet rejected. Testing stops when the entire test mass is allocated to non-rejected endpoints.

Figure 3 Multiple testing procedure



IDFS is planned to be analysed at the interim and the final analysis (see <u>Section 12.2.6</u> for further details). If IDFS is significant at the interim based on the ITT population then secondary endpoints will be formally tested at the interim based on the MTP outlined above. To account for multiple analyses on each endpoint a separate alpha spending function will be applied to each

NCI Version Date: 05-06-2021 142(177) NSABP B-55/BIG 6-13

endpoint (<u>Glimm et al 2010</u>). Further analyses of DDFS and OS with more mature follow up may be required for which some alpha will be reserved for significance testing.

# 12.2.6 Interim analysis

A superiority interim analysis of IDFS will occur when half the events needed for at least 90% power (165 events) have been observed from the first 50% of patients recruited (i.e. from first 900 patients) providing a cohort of patients with a similar level of maturity that is planned for the final analysis. Based on the database at time of amendment, the interim analysis is predicted to be October 2019 (80% CI: March 2019 to August 2020). The predictions will be tracked and monitored as more patients are enrolled in the study and additional data is added to the database. Two populations will be analysed at the interim analysis based on the analysis methods described in Section 12.2.1 for IDFS

- 1. Primary: ITT population (all patients randomised, estimated 254 events [80% CI: 226 to 289])
- 2. Supportive: Mature cohort population (first 900 patients randomised, 165 events anticipated)

The inclusion of a mature cohort population at the interim is to provide confidence that any observed treatment effect from the interim ITT population is maintained with longer-term follow-up. It is anticipated, based on the assumed recruitment and event rate that the interim analysis will occur approximately 5.3 years after the first patient is randomised and that all patients will have been randomised. At the time of the interim analysis, median time at risk per patient is expected to be 27 months in the ITT set, and 34 months in the mature cohort. The critical HR value at the interim analysis is 0.701.

Evidence of superiority for IDFS would only be determined at the interim if the results from both analysis populations provide evidence of a sustainable clinically relevant treatment effect for IDFS. More specifically, as a minimum the result in the ITT population would need to have met the statistical threshold defined below. Having met the statistical threshold in the ITT population, the result in the mature cohort (i.e. HR) would need to be of a similar magnitude such that the IDMC would consider it supportive of the ITT result and therefore have added confidence in the result in the ITT population. Statistical significance is not required for the mature cohort population. This analysis will be regarded as supportive, based on a cohort of patients with longer term follow-up, to aid interpretation of the result in the ITT population based on interim data. Other outcome measures such as 3 year IDFS rate will also be presented to aid the interpretation of the HRs (particularly in the case where the assumption of proportional hazards may not hold). KM plots will also be produced for IDFS.

The test mass alpha for IDFS (1 sided 2.5%) will be split between the final and the interim analysis using a bespoke spending function where a fixed significance level will be assigned at the interim and the remaining significance level assigned to the final analysis, taking account of correlation (Stone 2010). A 2-sided significance level of 0.005 will be assigned to the interim analysis so that a highly significant and clinically relevant result will need to be observed to declare superiority on IDFS. As an illustration, if 70% of the total required 330 IDFS events

NCI Version Date: 05-06-2021 143(177) NSABP B-55/BIG 6-13

have occurred in the ITT population at the interim then the observed HR would need to be < 0.7 for superiority to be declared. The HR in the mature cohort would need to be supportive of the ITT result. More detail around the criteria required for the mature cohort will be provided in the IDMC charter or SAP.

If the null hypothesis for IDFS is rejected at the interim for the ITT population then secondary endpoints (DDFS and OS) will be tested based on the MTP procedure outlined in <u>Section 12.2.5</u> using the significance levels provided in <u>Table 15</u>. If IDFS is not significant at the interim, DDFS and OS will not be tested at the IDFS interim and the significance level allocated to the IDFS interim for DDFS and OS will not be allocated to later timepoints.

Similar to IDFS, a bespoke spending function will be applied to the secondary endpoints OS and DDFS where a fixed significance level will be assigned to each analysis time point and the remaining significance level assigned to the final analysis time point controlling the overall type 1 error at the pre-specified alpha amount (Stone 2010). Provided the last analysis is known in advance of the penultimate one then the remaining alpha can be split to ensure that some alpha is always reserved for the final analysis. This approach allows flexibility in the number of analyses while appropriately controlling the overall type 1 error. Three analyses are planned for DDFS and four for OS for which some alpha will be reserved for significance testing. If additional analyses are required beyond the planned analyses and some alpha is still available for testing then any remaining alpha can be further split to strongly control the type 1 error (based on process described above). If no alpha remains then the additional analyses will be considered supportive updates of the already conducted analyses.

Given the split in alpha between DDFS and OS, if OS is significant based on the assigned significance level then the alpha assigned to OS will be recycled to DDFS and split across the planned analyses (and vice versa if DDFS is significant alpha for DDFS will be recycled to OS and split across analyses). The recycled alpha will be split based on the ratio of the originally assigned alpha split. For example if the original alpha allocation was split 1/3 for each analysis time point then the recycled alpha would also be split 1/3 across each analysis time point. For example, at the first interim analysis, assume IDFS is statistically significant and the secondary endpoint OS is also statistically significant. The significance level for testing DDFS is therefore 0.005 + (alpha assigned to OS recycled to DDFS and split across the planned analyses), i.e. <math>0.005 + (1% \* 0.005/0.04 = 0.00125) = 0.00625, or alternatively thought of as 0.005 \* 5/4.

Secondary endpoints will be assessed based on the ITT population. <u>Table 15</u> shows the different 2-sided significance levels that will be applied to the primary and secondary endpoints across the planned analyses as well as the total alpha spend for each endpoint. Note the significance level for the final analyses of each endpoint will be calculated using the relevant correlation based on the actual number of events for each analysis, the previous alpha spend and the total allocated alpha for that endpoint.

NCI Version Date: 05-06-2021 144(177) NSABP B-55/BIG 6-13

Table 15 Summary of 2-sided significance levels and total alpha spend across the endpoints and analyses

| | enupoints and | anaryses | | | |
|---|---|---|---|---|---|
| Endpoints | Interim<br>analysis | Final IDFS analysis | DDFS and OS analysis | Final OS analysis | |
| Estimated timings | | | | | |
| from FSI** | 5.3 years | 6.5 years | 10 years | 14 years | |
| | Significance<br>level | Significance level | Significance<br>level | Significance level | Total<br>alpha<br>spend (2-<br>sided) |
| IDFS | 0.005 | TBC* | N/A | N/A | 5% |
| If IDFS is stat<br>analysis | istically significant | and alpha is not recyc | eled between second | dary endpoints | at the |
| DDFS | 0.005 | 0.02 | TBC* | N/A | 4% |
| OS | 0.002 | 0.003 | 0.004 | TBC* | 1% |
| If IDFS is stat | istically significant | and alpha is recycled | between secondary | endpoints at th | e analysis |
| DDFS | 0.00625 | 0.025 | TBC* | N/A | 5% |
| OS | 0.01 | 0.015 | 0.02 | TBC* | 5% |

<sup>\*</sup>TBC: to be calculated; significance level to be calculated once relevant correlation based on the actual number of events for each analysis is known taking account of previous alpha spend and total allocated alpha \*\*FSI: first subject in

The IDMC will review the data from the interim analysis. The boundaries defined by the interim p-values for efficacy will be used as guidelines by the IDMC along with all other relevant trial information, including the safety data, to decide if it is appropriate to make a recommendation other than that to continue the trial as planned.

At the time of the interim analysis for superiority, an assessment of futility will also be performed. This futility assessment will be based on the probability of eventually showing statistical significance for the primary endpoint when the final number of IDFS events (n=330) is reached (<u>Lachin 2005</u>). The determination of this probability will be conditional on the observed data in the ITT population at the time of the interim analysis for superiority and on the assumed hazard ratio for the alternative hypothesis (IDFS HR=0.7). If the probability is less than 0.1, the IDMC will consider the option of declaring futility.

Full details on the process around the interim analysis and the efficacy criteria will be documented in the SAP and IDMC charter.

#### 12.2.7 Sample size justification

The primary endpoint of the study is IDFS and patients will be randomised 1:1 to either olaparib 300 mg b.i.d. (twice daily) or matching placebo.

NCI Version Date: 05-06-2021 145(177) NSABP B-55/BIG 6-13

A total of 1800 patients will be randomised into the study to achieve 330 IDFS events. If the true HR for the comparison of olaparib versus placebo in terms of IDFS is 0.7 then with 330 events, the analysis of IDFS will have 90% power to demonstrate a statistically significant difference in IDFS, assuming a 2-sided 5% significance level. The critical HR value at the primary analysis is 0.805.

The actual accrual pattern between June 2014 and February 2018 is shown in <u>Table 16</u>.

It is estimated that 1800 patients will be randomised by April/May 2019 so that the study will take approximately 5 years to complete recruitment (approximately 230 patients in US and approximately 1570 patients in the Rest of the World countries).

Table 16 Actual accrual between June 2014 and February 2018

| Interval since start of randomisation (months) | Number of patients randomized in interval | Cumulative number of patients randomized | Average number of patients randomized per month in interval |
|---|---|---|---|
| 0-6 | 21 | 21 | 3.5 |
| 6-12 | 94 | 115 | 15.7 |
| 12-18 | 174 | 289 | 29 |
| 18-24 | 180 | 469 | 33 |
| 24-30 | 229 | 698 | 38.2 |
| 30-36 | 249 | 947 | 41.5 |
| 36-42 | 234 | 1181 | 39 |
| 42-45* | 118 | 1299 | 39.3 |

<sup>\*</sup>Note: 3-month interval: December 2017 to February 2018 inclusive.

The primary analysis population will be all patients randomised (ITT). A subgroup analysis based on prior chemotherapy (adjuvant or neoadjuvant), prior platinum therapy (yes or no) and hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC) will be conducted to check for consistency in the treatment effect but this analysis is considered supportive of the primary analysis in the overall population.

During the trial, the Steering Committee will monitor the recruited patient population and actual event rate whilst remaining blinded to treatment. If the data suggests that the original sample size assumptions are incorrect such that achieving the required number of events with the current number of patients does not seem feasible then in consultation with the IDMC a decision may be made to increase the number of patients recruited into the trial to achieve the required 330 events.

NCI Version Date: 05-06-2021 146(177) NSABP B-55/BIG 6-13

#### 12.2.8 Issues relating to racial and ethnic differences in the U.S.

Possible racial and ethnic variation in response to the treatment under consideration is of great concern to. African-Americans. Researchers have noted poorer survival rates for African-American breast cancer patients as compared to Caucasians (<u>Baquet et al 1986</u>, <u>Youn et al 1984</u>). This difference has been attributed to many factors, including more advanced disease at the time of diagnosis (<u>Satariano et al 1986</u>), social and economic factors (<u>Bassett et al 1986</u>), or specific tumour characteristics such as ER positivity (<u>Crowe et al 1986</u>, <u>Mohla et al 1982</u>). Although outcomes tend to be less favorable for African-Americans, significant race-by-treatment interactions have not been previously reported suggesting that, where treatment efficacy exists, both groups appear to benefit. Previous NSABP investigations of the relationship between race and prognosis support these conclusions (<u>Dignam et al 1997</u>, <u>Costantino et al 1987</u>).

Potential for the enrolment of minority patients in this protocol is enhanced by the NRG Oncology's recognition of the importance of increasing minority accrual. To this end, we provide educational opportunities for NRG Oncology investigators and coordinators to increase their awareness and skills related to recruitment of racial and ethnic minority populations. The distributions of ethnicity and race for B-55/6-13 are projected from the NSABP B-40 study. The ethnicity distribution of the NSABP B-40 triple-negative population consists of 11% Hispanic and 89% non-Hispanic. The racial distribution in the triple-negative B-40 population is 84% white; 14% black, not of Hispanic origin; 1% Asian; < 1% Hawaiian or Pacific Islander descent; and < 1% American Indian or Alaskan Native.

The prognostic effect of race/ethnicity will be evaluated using statistical models. Unfortunately, because of power limitations, we will not be able to compare effects separately for the different cultural or racial groups.

Table 17 Expected racial and ethnic composition of NSABP B-55/BIG 6-13

| Ethnic Category | Total* |
|-------------------------------------------|--------|
| Hispanic or Latino | 25 |
| Not Hispanic or Latino | 205 |
| Ethnic Category: Total of all subjects | 230 |
| Racial Category | |
| American Indian or Alaskan Native | 1 |
| Asian | 2 |
| Black or African American | 32 |
| Native Hawaiian or other Pacific Islander | 2 |
| White | 193 |
| Racial Category: Total of all subjects | 230 |

<sup>\*</sup>Totals reflect the estimated accrual for U.S. sites only.

NCI Version Date: 05-06-2021 147(177) NSABP B-55/BIG 6-13
Ethnic Hispanic or Latino – a person of Cuban, Mexican, Puerto Rican, South or Categories: Central American, or other Spanish culture or origin, regardless of race.

**Not Hispanic or Latino** 

Racial Categories:

**American Indian or Alaskan Native** – a person having origins in any of the original peoples of North, Central or South America, and who maintains tribal affiliations or community attachment.

**Asian** – a person having origins in any of the original peoples of the Far East, Southeast Asia, or the Indian subcontinent including, for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, the Philippine Islands, Thailand, and Vietnam.

**Black or African American** – a person having origins in any of the black racial Groups of Africa.

Native Hawaiian or other Pacific Islander – a person having origins in any of the original peoples of Hawaii, Guam, Samoa, or other Pacific Islands.

**White** – a person having origins in any of the original peoples of Europe, the Middle East, or North Africa.

## 12.3 Independent data monitoring committee

This study will utilise an Independent Data Monitoring Committee (IDMC) whose members include therapeutic area experts and statisticians who are not employed by AstraZeneca and do not have any major conflict of interest. Members of the IDMC will be jointly selected by BIG, AstraZeneca, CTEP and NRG Oncology and the IDMC will report their recommendations to the Steering Committee.

The IDMC will meet approximately every 6 months and will review ongoing study progress including safety and, when appropriate, efficacy data. They will also review the data presented at the time of the protocol-defined interim analysis. The IDMC will have the ability to recommend suspension of enrolment if safety concerns are identified at any of the 6 monthly assessments. At the interim analysis both efficacy and safety will be reviewed and trial recommendations will be based on the totality of the data. The IDMC can recommend changes to the trial, including stopping of the trial, if they have concerns over the benefit risk profile for olaparib.

Reports for the IDMC will be prepared by an Independent Statistical Centre (ISC) and will be presented to the IDMC in closed session. Following review of data, the IDMC will make a recommendation regarding the future conduct of the trial to the Steering Committee. The IDMC recommendation will not contain any unblinded information or any information related to treatment outcomes of the trial.

A separate IDMC Charter will be developed defining the responsibilities and procedures for the IDMC.

NCI Version Date: 05-06-2021 148(177) NSABP B-55/BIG 6-13

## 13. IMPORTANT MEDICAL PROCEDURES TO BE FOLLOWED BY THE INVESTIGATOR

## 13.1 Medical emergencies and contacts

The Principal Investigator is responsible for ensuring that procedures and expertise are available to handle medical emergencies during the study. A medical emergency usually constitutes an SAE and is to be reported as such, see Section 6.4.10.

In the case of a medical emergency the investigator may contact the Protocol Officer. If the Protocol Officer is not available, contact one of the Protocol Chairs.

| Name | Role in the study | Address & telephone number |
|----------|-------------------|-------------------------------------|
| Redacted | Protocol Chair | Virginia Commonwealth<br>University |
| | | Redacted |
| Redacted | Protocol Chair | Dana-Farber Cancer Institute |
| | | Redacted |
| Redacted | Protocol Officer | NRG Oncology Redacted |

NCI Version Date: 05-06-2021 149(177) NSABP B-55/BIG 6-13

| Name | Role in the study | Address & telephone number |
|---|---|---|
| Redacted | Global Safety Physician | AstraZeneca |
| | | Redacted |
| | 24-hour emergency cover at NRG Oncology | Tel: Redacted |
| For routine clinical questions, contact the Clinical Coordinating Department: | | |
| Redacted | | |

### 13.2 Overdose

There is currently no specific treatment in the event of overdose with olaparib and possible symptoms of overdose are not established. Study treatment must only be used in accordance with the dosing recommendations in this protocol. Any dose or frequency of dosing that exceeds the dosing regimen specified in this protocol should be reported as an overdose. Any overdose should be reported as a minor protocol deviation. The MTD is 300 mg b.i.d (tablet).

Adverse reactions associated with overdose should be treated symptomatically and should be managed appropriately.

- An overdose with associated AEs is recorded as the AE diagnosis/symptoms on the relevant AE modules in the eCRF and on the Overdose eCRF module.
- An overdose without associated symptoms is only reported on the Overdose eCRF module.

If an overdose on an AstraZeneca study drug occurs in the course of the study, then Investigators or other site personnel inform the Protocol Officer immediately, or no later than 24 hours of when he or she becomes aware of it.

The Protocol Officer works with the Investigator to ensure that all relevant information is provided to NRG Oncology.

For overdoses associated with SAE, standard reporting timelines apply (see <u>Section 6.4.10</u>). For other overdoses, reporting should be done within 30 days.

## 13.3 Pregnancy

All outcomes of pregnancy should be reported via CTEP-AERS.

## 13.3.1 Maternal exposure

If a patient becomes pregnant during the course of the study the investigational product should be discontinued immediately. Call the NRG Oncology Clinical Coordinating Department (see <u>Information Resources</u>).

NCI Version Date: 05-06-2021 150(177) NSABP B-55/BIG 6-13

The outcomes of any conception occurring from the date of the first dose of study medication until 3 months after the last dose of study medication must be followed up and documented.

Pregnancy itself is not regarded as an adverse event unless there is a suspicion that the investigational product under study may have interfered with the effectiveness of a contraceptive medication. Congenital abnormalities/birth defects and spontaneous miscarriages should be reported and handled as SAEs. Elective abortions without complications should not be handled as AEs. The outcome of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal birth or congenital abnormality) should be followed up and documented even if the patient was discontinued from the study medication.

## 13.3.2 Expedited reporting of pregnancy, pregnancy loss, and death neonatal occurring during study therapy

Any pregnancy, pregnancy loss, or death neonatal occurring while the patient is receiving study therapy or within 3 months following the last dose of study therapy must be reported via CTEP-AERS as a medically significant event. Definitions and reporting instruction for these events are provided in the Cancer Therapy Evaluation Program's (CTEP) revised NCI guidelines for Investigators: Adverse Event Reporting Requirements (Section 5.5.6) located at the following CTEP website:

 $(\underline{http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/aeguidelines.pdf}).$ 

Upon learning of a pregnancy, pregnancy loss, or death neonatal that occurs during study or within 3 months following the last dose of study therapy the investigator is required to:

- Within 5 working days of learning of the event, and as required by the NCI Guidelines for Investigators: Adverse Event Reporting Requirements (Section 5.5.6):
  - Create and submit a CTEP-AERS report;
  - Complete the Pregnancy Information Form (located on the CTEP website at http://ctep.cancer.gov/protocolDevelopment/adverse effects.htm); and
  - Fax the completed Pregnancy Information Form with all available supporting documentation to the NRG Oncology SDMC's expedited fax number at 412-622-2113.
- The pregnancy outcome for patients on study should be reported via CTEP-AERS at the time the outcome becomes known, accompanied by the same Pregnancy Information Form used for the initial report.
- For questions concerning AE reporting, contact the AE Reporting Nurse (see <u>Information</u> Resources).

## 13.3.3 Paternal exposure

Male patients should refrain from fathering a child or donating sperm during the study treatment period and for 3 months following the last dose. Pregnancy of the patient's partners is not considered to be an adverse event. However, the outcome of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal birth or congenital abnormality) should if possible be followed up and documented.

The outcome of any conception occurring from the date of the first dose until 3 months after the last dose should be followed up and documented.

NCI Version Date: 05-06-2021 151(177) NSABP B-55/BIG 6-13

#### 14. LIST OF REFERENCES

#### Aaronson et al 1993

Aaronson NK, Ahmedzai S, Bergman B, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst 1993; 85(5):365-376.

#### Aebi et al 2011

S. Aebi, T. Davidson, G. Gruber & F. Cardoso. Primary breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Annals of Oncology 22 (Supplement 6): vi12–vi24, 2011.

## **American Cancer Society 2013**

American Cancer Society. Cancer Facts and Figures 2013. Atlanta, Georgia: American Cancer Society, 2013. http://www.cancer.org.

#### Antoniou et al 2003

Antoniou A, Pharoah PD, Narod S, Risch HA, Eyfjord JE, Hopper JL, et al. Average risks of breast and ovarian cancer associated with *BRCA*1 or *BRCA*2 mutations detected in case Series unselected for family history: a combined analysis of 22 studies. Am J Hum Genet 2003;72(5):1117-30.

#### Arun et al 2011

Arun B, Bayraktar S, Liu DD, Gutierrez Barrera AM, Atchley D, Pusztai L, et al. Response to neoadjuvant systemic therapy for breast cancer in *BRCA* mutation carriers and non-carriers: a single-institution experience. J Clin Oncol 2011; 29(28):3739-46.

#### Atchley et al 2008

Atchley DP, Albarracin CT, Lopez A, Valero V, Amos CI, Gonzalez-Angulo AM, et al. Clinical and pathologic characteristics of patients with *BRCA*-positive and *BRCA*-negative breast cancer. J Clin Oncol. 2008; 26(26):4282-8.

#### Baquet et al 1986

Baquet CR, Ringen K, Pollack ES, et al. Cancer Among Blacks and Other Minorities: Statistical Profiles. Bethesda MD: National Institutes of Health. DHEW publication (NIH), 1986; 86:2785.

#### Bassett et al 1986

Bassett MT, Krieger N. Social class and black-white differences in breast cancer survival. Am J Public Health 1986; 76:1400-1403.

#### Bergfeldt et al 1995

Bergfeldt K, Einhorn S, Rosendahl I, Hall P. Increased risk of second primary malignancies in patients with gynecological cancer. A Swedish record-linkage study. Acta Oncol. 1995;34(6):771-7.

NCI Version Date: 05-06-2021 152(177) NSABP B-55/BIG 6-13

#### Bernhard J et al 2007

Bernhard J, Zahrieh D, Castiglione-Gertsch M, et al. Adjuvant chemotherapy followed by goserelin compared with either modality alone: the impact on amenorrhea, hot flashes, and quality of life in premenopausal patients—the International Breast Cancer Study Group Trial VIII. J Clin Oncol 2007; 25:263-270.

#### Bordeleau et al 2011

Bordeleau L, Lipscombe L, Lubinski J, et al. Diabetes and breast cancer among women with *BRCA*1 and *BRCA*2 mutations. Cancer 2011;117:1812-8.

#### Bower et al 2000

Bower JE, Ganz PA, Desmond KA, et al. Fatigue in breast cancer survivors: occurrence, correlates, and impact on quality of life. J Clin Oncol 2000; 18(4):743-753.

#### Bower et al 2006

Bower JE, Ganz PA, Desmond KA, et al. Fatigue in long-term breast carcinoma survivors: a longitudinal investigation. Cancer 2006; 106(4):751-758.

#### Burnell et al 2010

Burnell M, Levine MN, Chapman JW, Bramwell V, Gelmon K, Walley B, et al. Cyclophosphamide, Epirubicin, and Fluorouracil Versus Dose-Dense Epirubicin and Cyclophosphamide Followed by Paclitaxel Versus Doxorubicin and Cyclophosphamide Followed by Paclitaxel in Node-Positive or High-Risk Node-Negative Breast Cancer. Journal of Clinical Oncology;vol28 no 1.

## Cameron et al 2013

Cameron D, Brown J, Dent R et al. Adjuvant bevacizumab-containing therapy in triple-negative breast cancer (BEATRICE): primary results of a randomised, phase 3 trial. Lancet Oncol 2013; 14:933-42.

## **Carey 2011**

Carey LA. Directed Therapy of Subtypes of Triple-Negative Breast Cancer. The Oncologist 2011;16(suppl 1):71–78.

#### Cella D et al 2002

Cella D, Eton DT, Lai JS, et al. Combining anchor and distribution-based methods to derive minimal clinically important differences on the Functional Assessment of Cancer Therapy (FACT) anemia and fatigue scales. J Pain Symptom Manage 2002; 24(6):547-561

### **Cole and Strair 2010**

Cole M, Strair R. Acute myelogenous leukemia and myelodysplasia secondary to breast cancer treatment: case studies and literature review. Am J Med Sci 2010;339(1):36-40.

#### Cortazar et al 2014

Cortazar P, Zhang L, Untch M, et al. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet 2014; 384:164-72.

NCI Version Date: 05-06-2021 153(177) NSABP B-55/BIG 6-13

#### Costantino et al 1987

Costantino JP, Redmond CK, Wickerham D, et al. A comparison of survival between white and black breast cancer patients: Results from NSABP B-09. Proc Am Soc Clin Oncol 1987; 6:230 Abstr 905.

#### Crowe et al 1986

Crowe JP Jr, Gordon NH, Hubay CA, et al. The interaction of estrogen receptor status and race in predicating prognosis for stage I breast cancer patients. Surgery 1986; 100:599-605.

#### Dent et al 2007

Dent R, Trudeau M, Pritchard KI, Hanna WM, Kahn HK, Sawka CA, Lickley LA, Rawlinson E, Sun P, Narod SA. Triple-negative breast cancer: clinical features and patterns of recurrence. Clin Cancer Res. 2007;13:4429-34.

#### Dignam et al 1997

Dignam JJ, Redmond CK, Fisher B, et al. Prognosis among African-American women and white women with lymph node-negative breast carcinoma: Findings from two randomized clinical trials of the National Surgical Adjuvant Breast and Bowel Project (NSABP). Cancer 1997; 80:80-90.

## Fine and Gray 1999

Fine, J. and Gray, R. A proportional hazards model for the subdistribution of a competing risk. Journal of the American Statistical Association 1999;94,496-509.

## Fong et al 2009

Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, et al. Inhibition of poly(ADPribose) polymerase in tumors from *BRCA* mutation carriers. N Engl J Med. 2009;361(2);123-34.

## Foulkes et al 2010

Foulkes, W, Smith, IE, Reis-Filho, JS. Triple Negative Breast Cancer. N Engl J Med 2010;363;1938-48.

#### Fowble et al 2001

Fowble B, Hanlon A, Freedman G, Nocolaou N, Anderson P. Second cancers after conservative surgery and radiation for stages I-II breast cancer: identifying a subset of women at increased risk. Int J Radiat Oncol, Biol, Phys. 2001; 51 (3):679-690.

#### Gail and Simon 1985

Gail M, Simon R. Testing for qualitative interactions between treatment effects and patient subsets. Biometrics 1985;41:361-72.

#### Ganz et al 1998A

Ganz PA, Rowland JH, Desmond K, et al. Life after breast cancer: understanding women's health-related quality of life and sexual functioning. J Clin Oncol 1998; 16(2):501-514.

NCI Version Date: 05-06-2021 154(177) NSABP B-55/BIG 6-13

#### Ganz et al 1998B

Ganz PA, Rowland JH, Meyerowitz BE, et al. Impact of different adjuvant therapy strategies on quality of life in breast cancer survivors. Recent Results Cancer Res 1998; 152(9):396-411.

#### Ganz et al 2002

Ganz PA, Desmond KA, Leedham B, et al. Quality of life in long-term, disease-free survivors of breast cancer: a follow-up study. J Natl Cancer Inst 2002; 94(1):39-49.

#### Ganz et al 2004

Ganz PA, Kwan L, Stanton AL, et al. Quality of life at the end of primary treatment of breast cancer: first results from the moving beyond cancer randomized trial. J Natl Cancer Inst 2004; 96(5):376-387.

#### Ganz et al 2011A

Ganz PA, Kwan L, Stanton AL, et al. Physical and psychosocial recovery in the year after primary treatment of breast cancer. J Clin Oncol 2011; 29(9):1101-1109.

#### Ganz et al 2011B

Ganz PA, Land SR, Geyer CE, et al. Menstrual history and quality-of-life outcomes in women with node-positive breast cancer treated with adjuvant therapy on the NSABP B-30 trial. J Clin Oncol 2011; 29(9):1110-1116.

#### Gaymes et al 2008

Gaymes TJ, Shall S, MacPherson LJ, Twine NA, Lea NC, Farzaneh F, and Mufti GJ. Inhibitors of poly ADP-ribose polymerase (PARP) induce apoptosis of myeloid leukemic cells: potential for therapy of myeloid leukemia and myelodysplastic syndromes. Haematologica 2009; 94:638-646. doi:10.3324/haematol.2008.001933.

#### Gelmon et al 2011

Gelmon KA, Tischkowitz M, Mackay H, Swenerton K, Robidoux A, Tonkin K, et al. Olaparib in patients with recurrent high-grade serous or poorly differentiated ovarian carcinoma or triplenegative breast cancer: a phase 2, multicentre, open-label, non-randomised study. Lancet Oncol 2011; 12: 852–61

#### Ginsburg et al 2010

Ginsburg OM, Kim-Sing C, Foulkes WD, Ghadirian P, Lynch HT, Sun P, et al. *BRCA*1 and *BRCA*2 families and the risk of skin cancer. Fam Cancer 2010; 9:489-93.

#### Glimm et al 2010

Glimm, E., Maurer, W., and Bretz, F. Hierarchical testing of multiple endpoints in group-sequential trials. Statistics in Medicine 2010;29, 219–228.

#### Goodwin et al 2012

Goodwin PJ, Phillips KA, West DW, et al. Breast cancer prognosis in *BRCA*1 and *BRCA*2 mutation carriers: An international perspective breast cancer family registry population-based cohort study. J Clin Oncol 2012;30:19-26.

NCI Version Date: 05-06-2021 155(177) NSABP B-55/BIG 6-13

### Gupta et al 2007

Gupta B, Sait SN, Block AW, Ford LA, moysich KB, Baer MR. Acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) following treatment for ovarian cancer. J Clin Oncol 2007;ASCO Annual Meeting Proceedings Part 1,Vol 25, No 18S:17506.

## Hay et al 2009

Hay T, Matthews JR, Pietzka L, Lau A, Cranston A, Nygren AO, et al. Poly(ADP-ribose) polymerase-1 inhibitor treatment regresses autochthonous *BRCA* 2/p53-mutant mammary tumors in vivo and delays tumor relapse in combination with carboplatin. Cancer Res. 2009;69(9):3850-5.

## Helleday 2011

Helleday T. The underlying mechanism for the PARP and *BRCA* synthetic lethality: Clearing up the misunderstandings. Molecular Oncology 2011; 5: 387-393.

#### Hershman et al 2007

Hershman D, Neugut AI, Jacobson JS, Wang J, Tsai W, McBride R, Bennett CL, Grann VR. Acute Myeloid Leukemia or Myelodysplastic Syndrome Following Use of Granulocyte Colony-Stimulating Factors During Breast Cancer Adjuvant Chemotherapy. JNCI 2007 Vol. 99, Issue 3,Febr7.

## Honrado et al 2006

Honrado E, Benítez J, Palacios J. Histopathology of *BRCA*1- and *BRCA*2-associated breast cancer. Crit Rev Oncol Hematol 2006; 59:27-39.

## Hudis et al 2007

Hudis CA, William E, Barlow JP, Costantino RJ, Gray KI, Pritchard J-AW, et al. Proposal for Standardized Definitions for Efficacy End Points in Adjuvant Breast Cancer Trials: The STEEP System. J Clin Oncol 2007;25(15):2127-32.

#### Huzarski et al 2013

Huzarski T, Byrski T et al. Ten-Year Survival in Patients With *BRCA*1-Negative and *BRCA*1-Positive Breast Cancer. J Clin Oncol 2013; 31:3191-3196.

#### Jeruss et al 2008

Jeruss SJ, Mittendorf EA et al. Combined Use of Clinical and Pathologic Staging Variables to Define Outcomes for Breast Cancer Patients Treated With Neoadjuvant Therapy. J Clin Oncol 2008; J Clin Oncol 26:246-252.

#### Kaufman et al 2014

Kaufman B, Shapira-Frommer R et al. Olaparib monotherapy in patients with advanced cancer and a germline *BRCA1/2* mutation. J Clin Oncol 2014 Nov 3.pii: JCO.2014.56.2728.

## Khatcheressian et al 2012

Khatcheressian JL, Hurley P et al. Breast Cancer Follow-Up and Management after primary treatment: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol 30, 2012.

NCI Version Date: 05-06-2021 156(177) NSABP B-55/BIG 6-13

#### Lachin 2005

Lachin, J. M. (2005). A review of methods for futility stopping based on conditional power. Statist. Med., 24: 2747–2764. Statist Med 24:2747-2764

#### Liedtke et al 2008

Liedtke, C, Mazouni C, Hess K, Andre' F, Tordai A, Mejia JA, et al. Response to Neoadjuvant Therapy and Long-Term Survival in Patients With Triple-Negative Breast Cancer. J Clin Oncol 2008; 26(8).

#### Mavaddat et al 2012

Mavaddat et al. Pathology of breast and ovarian cancers among *BRCA*1 and *BRCA*2 mutation carriers: results from the Consortium of Investigators of Modifiers of *BRCA*1/2 (CIMBA) Cancer Epidemiol Biomarkers Prev. 2012 January; 21(1): 134–147. doi:10.1158/1055-9965.EPI-11-0775.

## Metzger-Filho et al 2010

Metzger-Filho O, Tutt A, de Azambuja E, Saini KS, Viale G, Loi S, et al. Disecting the heterogeneity of triple negative breast cancer. J Clin Oncol. 2012 May 20;30 915:1879-87. Doi: 10.1200/JCO.2011.38.2010.

#### Mieog et al 2007

Mieog JS, van der Hage JA, van de Velde CJ. Preoperative chemotherapy for women with operable breast cancer. Cochrane Database Syst Rev. 2007;18(2):CD005002.

#### Mittendorf et al 2011

Mittendorf EA, Jeruss JS, Tucker SL, Kolli A, Newman LA, Gonzalez-Angulo et al. Validation of a Novel Staging System for Disease-Specific Survival in Patients With Breast Cancer Treated With Neoadjuvant Chemotherapy. Journal of Clinical Oncology 2011 vol 29 no 15 may.

#### Mohla et al 1982

Mohla S, Sampson CC, Khan T, et al. Estrogen and progesterone receptors in breast cancer in black Americans: Correlation of receptor data with tumor differentiation. Cancer 1982; 50:552-559.

#### Morton et al 2013

Morton LM, Dores GM, Tucker MA, Kim CJ, Onel K, Gilbert ES, et al. Evolving risk of therapy-related acute myeloid leukemia following cancer chemotherapy among adults in the United States, 1975-2008. Blood 2013;121(15):2996-3004.

#### Murai et al 2012

Murai J, Huang SN, Das BB, Renaud A, et al. Trapping of PARP1 and PARP2 by Clinical PARP Inhibitors. AACR 2012; 72(21); 5588–99.

#### Nardone et al 2015

Nardone A, Goldstein A, Shea MJ, Mithchell T, Fu X, De C et al. PARP inhibition effects on endocrine therapy and resistance in estrogen receptor positive (ER+) breast cancer models. AACR 2015, abstract # 15LB8846AACR.

NCI Version Date: 05-06-2021 157(177) NSABP B-55/BIG 6-13

#### Praga et al 2005

Praga C, Bergh J, Bliss J, Bonneterre J, Cesana B, Coombes RC, et al. Risk of Acute Myeloid Leukemia and Myelodysplastic Syndrome in Trials of Adjuvant Epirubicin for Early Breast Cancer: Correlation With Doses of Epirubicin and Cyclophosphamide. J Clinl Oncol 2005; 23(18):4179-4191.

#### Rennert et al 2007

Rennert G, Bisland-Naggan S, Barnett-Griness O, Bar-Joseph N, Zhang S, Hedy S. Clinical outcomes of breast cancer in carriers of *BRCA*1 and *BRCA*2 mutations. N Engl J Med 2007;357:115-23.

### Rottenberg et al 2008

Rottenberg S, Jaspers JE, Kersbergen A, van der Burg E, Nygren AO, Zander SA, et al. High sensitivity of *BRCA*1-deficient mammary tumors to the PARP inhibitor AZD2281 alone and in combination with platinum drugs. Proc Natl Acad Sci. 2008;105(44):17079-84.

#### Robins et al 1991

Robins JM, Tsiatis AA. Correcting for noncompliance in randomized trials using rank preserving structural failure time models. Communications in Statistics - Theory and Methods 1991; 20:2609-2631.

#### Robson et al 2004

Robson ME, Chappuis PO, Satagopan J, Wong N, Boyd J, Goffin JR, et al. A combined analysis of outcome following breast cancer: Differences in survival based on *BRCA1/BRCA2* mutation status and administration of adjuvant treatment. Breast Cancer Res 2004;6(1):R8-17.

## Robson et al 2017

Robson M, Im SA, Senkus E, Xu B, Domchek SM, Masuda N, et al. Olaparib for metastatic breast cancer in patients with a germline BRCA mutation. N Engl J Med 2017;377(6):522-33.

### Satariano et al 1986

Satariano WA, Belle SH, Swanson GM. The severity of breast cancer at diagnosis: A comparison of age and extent of disease in black and white women. Am J Public Health 1986; 76:779-782.

## Schiewer et al 2013

Schiewer MJ, Goodwin JF, Han S, Brenner JC, Augello MA, Dean JL, et al. Dual roles of PARP-1 promote cancer growth and progression. Cancer Discov. 2012;2(12):1134-49.

## Smith et al 2003

Smith RE, Bryant J, DeCillis A, Anderson S. Acute Myeloid Leukemia and Myelodysplastic Syndrome After Doxorubicin-Cyclophosphamide Adjuvant Therapy for Operable Breast Cancer: The National Surgical Adjuvant Breast and Bowel Project Experience 2003 J Clin Oncol 21:1195-1204.

NCI Version Date: 05-06-2021 158(177) NSABP B-55/BIG 6-13

#### **Stone 2010**

A Stone. The application of bespoke spending functions in group-sequential designs and the effect of delayed treatment switching in survival trials. Pharmaceutical statistics 2010; 9, 151-161

#### Swain et al 2013

Swain SM, Tang G, Geyer CE Jr, Rastogi P, Atkins JN, Donnellan PP, et al. Definitive results of a phase III adjuvant trial comparing three chemotherapy regimens in women with operable, node-positive breast cancer: the NSABP B-38 trial. J Clin Oncol. 2013 Sep 10;31(26):3197-204.

## Tryggvadottir et al 2013

Tryggvadottir L, Olafsdottir EJ, Olafsdottir GH, Sigurdsson H, Johannsson OT, Bjorgvinsson E, et al. Tumour diploidy and survival in breast cancer patients with BRCA2 mutations. Breast Cancer Res Treat 2013 Jul;140:375–38.

#### Tutt et al 2010

Tutt A, Robson M, Garber JE, Domchek SM, Audeh MW, Weitzel JN, et al. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with *BRCA*1 or *BRCA*2 mutations and advanced breast cancer: a proof-of-concept trial. Lancet 2010; 376: 235–44.

#### **Vay et al 2011**

Vay A, Kumar S, Seward S, Semaan A, Schiffer CA, Munkarah AR at al. Therapy-related myeloid leukemia after treatment for epithelial ovarian carcinoma: an epidemiological analysis. Gynecologic Oncology 2011;123:456-60.

#### Von Minckwitz et al 2012

Von Minckwitz G, Untch M, Blohmer JU et al. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol 2012; 30: 1796–1804.

#### Wesolowski et al 2007

Wesolowski R, Choueiri TK, Rybicki L, Shealy AG, Casey G, Weng D, et al. *BRCA* mutation status and risk of secondary malignancy following chemotherapy for breast cancer. J Clin Oncol, 2007;ASCO Annual Meeting Proceedings Part I. Vol (25);No. 18S (June 20 Supplement):11017.

#### Yellen et al 1997

Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemiarelated symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage 1997; 13(2), 63-74.

## Youn et al 1984

Youn JL Jr, Ries LG, Pollack ES. Cancer patient survival among ethnic groups in the United States. J Natl Cancer Inst 1984; 73:341-352.

## Zhang et al 2013

Zhang F, Wang Y, Wang L, Luo X, Huang K, Wang C, Du M, Liu F, Luo T, Huang D, Huang K. Poly(ADP-ribose) polymerase 1 is a key regulator of estrogen receptor α-dependent gene transcription. J Biol Chem. 2013;288(16):11348-57.

NCI Version Date: 05-06-2021 159(177) NSABP B-55/BIG 6-13

## **Appendix A** Additional Safety Information

## Further Guidance on the Definition of a Serious Adverse Event (SAE)

## Life threatening

'Life-threatening' means that the subject was at immediate risk of death from the AE as it occurred or it is suspected that use or continued use of the product would result in the subject's death. 'Life-threatening' does not mean that had an AE occurred in a more severe form it might have caused death (e.g., hepatitis that resolved without hepatic failure).

#### Hospitalisation

Outsubject treatment in an emergency room is not in itself a serious AE, although the reasons for it may be (e.g., bronchospasm, laryngeal oedema). Hospital admissions and/or surgical operations planned before or during a study are not considered AEs if the illness or disease existed before the subject was enrolled in the study, provided that it did not deteriorate in an unexpected way during the study.

### Important medical event or medical intervention

Medical and scientific judgement should be exercised in deciding whether a case is serious in situations where important medical events may not be immediately life threatening or result in death, hospitalisation, disability or incapacity but may jeopardize the subject or may require medical intervention to prevent one or more outcomes listed in the definition of serious. These should usually be considered as serious.

Simply stopping the suspect drug does not mean that it is an important medical event; medical judgement must be used.

## Examples of such events are:

- Angioedema not severe enough to require intubation but requiring iv hydrocortisone treatment
- Hepatotoxicity caused by paracetamol (acetaminophen) overdose requiring treatment with N-acetylcysteine
- Intensive treatment in an emergency room or at home for allergic bronchospasm
- Blood dyscrasias (e.g., neutropenia or anaemia requiring blood transfusion, etc) or convulsions that do not result in hospitalisation
- Development of drug dependency or drug abuse.

NCI Version Date: 05-06-2021 160(177) NSABP B-55/BIG 6-13

## A Guide to Interpreting the Causality Question

The following factors should be considered when deciding if there is a "reasonable possibility" that an AE may have been caused by the drug.

- Time Course. Exposure to suspect drug. Has the subject actually received the suspect drug? Did the AE occur in a reasonable temporal relationship to the administration of the suspect drug?
- Consistency with known drug profile. Was the AE consistent with the previous knowledge of the suspect drug (pharmacology and toxicology) or drugs of the same pharmacological class? OR could the AE be anticipated from its pharmacological properties?
- Dechallenge experience. Did the AE resolve or improve on stopping or reducing the dose of the suspect drug?
- No alternative cause. The AE cannot be reasonably explained by another aetiology such as the underlying disease, other drugs, other host or environmental factors.
- Rechallenge experience. Did the AE reoccur if the suspected drug was reintroduced after having been stopped? AstraZeneca would not normally recommend or support a rechallenge.
- Laboratory tests. A specific laboratory investigation (if performed) has confirmed the relationship?

A "reasonable possibility" could be considered to exist for an AE where one or more of these factors exist.

In contrast, there would not be a "reasonable possibility" of causality if none of the above criteria apply or where there is evidence of exposure and a reasonable time course but any dechallenge (if performed) is negative or ambiguous or there is another more likely cause of the AE.

In difficult cases, other factors could be considered such as:

- Is this a recognised feature of overdose of the drug?
- Is there a known mechanism?

Ambiguous cases should be considered as being a "reasonable possibility" of a causal relationship unless further evidence becomes available to refute this. Causal relationship in cases where the disease under study has deteriorated due to lack of effect should be classified as no reasonable possibility.

NCI Version Date: 05-06-2021 161(177) NSABP B-55/BIG 6-13

# **Appendix B** International Airline Transportation Association (IATA) 6.2 Guidance Document

## **Labelling and Shipment of Biohazard Samples**

International Airline Transportation Association (IATA) classifies biohazardous agents into 3 categories. For transport purposes the classification of infectious substances according to risk groups was removed from the Dangerous Goods Regulations (DGR) in the 46th edition (2005). Infectious substances are now classified either as Category A, Category B or Exempt. There is no direct relationship between Risk Groups and categories A and B.

Category A Infectious Substances are infectious substances in a form that, when exposure to it occurs, is capable of causing permanent disability, life-threatening or fatal disease in otherwise healthy humans or animals. Category A pathogens are e.g., Ebola, Lassa fever virus:

• are to be packed and shipped in accordance with IATA Instruction 602.

**Category B Infectious Substances** are infectious Substances that do not meet the criteria for inclusion in Category A. Category B pathogens are e.g., Hepatitis A, B, C, D, and E viruses, Human immunodeficiency virus (HIV) types 1 and 2. They are assigned the following UN number and proper shipping name:

- UN 3373 Biological Substance, Category B
- are to be packed in accordance with UN3373 and IATA 650

**Exempt** - all other materials with minimal risk of containing pathogens

- Clinical trial samples will fall into Category B or exempt under IATA regulations
- Clinical trial samples will routinely be packed and transported at ambient temperature in IATA 650 compliant packaging
- Biological samples transported in dry ice require additional dangerous goods specification for the dry-ice content
- IATA compliant courier and packaging materials should be used for packing and transportation and packing should be done by an IATA certified person, as applicable
- Samples routinely transported by road or rail are subject to local regulations which require that they are also packed and transported in a safe and appropriate way to contain any risk of infection or contamination by using approved couriers and packaging / containment materials at all times. The IATA 650 biological sample containment standards are encouraged wherever possible when road or rail transport is used.

NCI Version Date: 05-06-2021 162(177) NSABP B-55/BIG 6-13









# Appendix D Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law

#### Introduction

This Appendix describes the process to be followed in order to identify and appropriately report cases of Hy's Law. It is not intended to be a comprehensive guide to the management of elevated liver biochemistries.

During the course of the study the Investigator will remain vigilant for increases in liver biochemistry. The investigator is responsible for determining whether a subject meets potential Hy's Law (PHL) criteria at any point during the study.

The Investigator participates, together with the Protocol Officer, in review and assessment of cases meeting PHL criteria to agree whether Hy's Law (HL) criteria are met. HL criteria are met if there is no alternative explanation for the elevations in liver biochemistry other than Drug Induced Liver Injury (DILI) caused by the Investigational Medicinal Product (IMP).

The Investigator is responsible for recording data pertaining to PHL/HL cases and for reporting Adverse Events (AE) and Serious Adverse Events (SAE) according to the outcome of the review and assessment in line with standard safety reporting processes.

#### **Definitions**

### Potential Hy's Law (PHL)

Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)  $\geq$  3x Upper Limit of Normal (ULN) **together with** Total Bilirubin (TBL)  $\geq$  2xULN at any point during the study following the start of study medication irrespective of an increase in Alkaline Phosphatase (ALP).

### Hy's Law (HL)

AST or ALT  $\geq$  3x ULN **together with** TBL  $\geq$  2xULN, where no other reason, other than the IMP, can be found to explain the combination of increases, e.g., elevated ALP indicating cholestasis, viral hepatitis, another drug.

For PHL and HL the elevation in transaminases must precede or be coincident with (i.e. on the same day) the elevation in TBL, but there is no specified timeframe within which the elevations in transaminases and TBL must occur.

## **Identification of Potential Hy's Law Cases**

In order to identify cases of PHL it is important to perform a comprehensive review of laboratory data for any subject who meets any of the following identification criteria in isolation or in combination:

• ALT  $\geq 3xULN$ 

NCI Version Date: 05-06-2021 167(177) NSABP B-55/BIG 6-13

- AST  $\geq 3xULN$
- TBL  $\geq 2xULN$

The Investigator will without delay review each new laboratory report and if the identification criteria are met will:

- Determine whether the subject meets PHL criteria (see <u>Definitions</u> within this Appendix for definition) by reviewing laboratory reports from all previous visits
- Promptly enter the laboratory data into the laboratory CRF

#### Follow-Up

## Potential Hy's Law Criteria not met

If the subject does not meet PHL criteria the Investigator will:

• Perform follow-up on subsequent laboratory results according to the guidance provided in the Clinical Study Protocol.

## Potential Hy's Law Criteria met

If the subject does meet PHL criteria the Investigator will:

• Notify the Protocol Officer

The Protocol Officer contacts the Investigator, to provide guidance, discuss and agree an approach for the study subjects' follow-up and the continuous review of data. Subsequent to this contact the Investigator will:

- Monitor the subject until liver biochemistry parameters and appropriate clinical symptoms and signs return to normal or baseline levels, or as long as medically indicated
- Investigate the etiology of the event and perform diagnostic investigations as discussed with the Study Physician
- Complete the three Liver CRF Modules as information becomes available
- If at any time (in consultation with the Protocol Officer) the PHL case meets serious criteria, report it as an SAE using standard reporting procedures

#### Review and Assessment of Potential Hy's Law Cases

The instructions in this Section should be followed for all cases where PHL criteria are met.

No later than 3 weeks after the biochemistry abnormality was initially detected, the Protocol Officer contacts the Investigator in order to review available data and agree on whether there is an alternative explanation for meeting PHL criteria other than DILI caused by the IMP. The AstraZeneca Medical Science Director and Global Safety Physician will also be involved in this review together with other subject matter experts as appropriate.

According to the outcome of the review and assessment, the Investigator will follow the instructions below.

If there **is** an agreed alternative explanation for the ALT or AST and TBL elevations, a determination of whether the alternative explanation is an AE will be made and subsequently whether the AE meets the criteria for a SAE:

- If the alternative explanation is **not** an AE, record the alternative explanation on the appropriate CRF
- If the alternative explanation is an AE/SAE, record the AE /SAE in the CRF accordingly and submit (see <u>Sections 6.4.9</u> and <u>6.4.10</u> of the protocol)

If it is agreed that there is **no** explanation that would explain the ALT or AST and TBL elevations other than the IMP:

- Report an SAE (report term 'Hy's Law') via CTEP-AERS.
  - The 'Medically Important' serious criterion should be used if no other serious criteria apply
  - As there is no alternative explanation for the HL case, a causality assessment of 'related' should be assigned.

If, there is an unavoidable delay, of over 3 weeks, in obtaining the information necessary to assess whether or not the case meets the criteria for HL, then it is assumed that there is no alternative explanation until such time as an informed decision can be made:

- Report an SAE (report term 'Potential Hy's Law') applying serious criteria and causality assessment as per above
- Continue follow-up and review according to agreed plan. Once the necessary supplementary information is obtained, repeat the review and assessment to determine whether HL criteria are met. Update the SAE report according to the outcome of the review amending the reported term if an alternative explanation for the liver biochemistry elevations is determined.

NCI Version Date: 05-06-2021 169(177) NSABP B-55/BIG 6-13

## Actions Required for Repeat Episodes of Potential Hy's Law

This section is applicable when a subject meets PHL criteria on study treatment and has already met PHL criteria at a previous on study treatment visit.

The requirement to conduct follow-up, review and assessment of a repeat occurrence(s) of PHL is based on the nature of the alternative cause identified for the previous occurrence.

The investigator should determine the cause for the previous occurrence of PHL criteria being met and answer the following question:

• Was the alternative cause for the previous occurrence of PHL criteria being met found to be the disease under study e.g. chronic or progressing malignant disease, severe infection or liver disease?

If No: follow the process described in Potential Hy's Law Criteria met of this Appendix

#### If Yes:

Determine if there has been a significant change in the subject's condition<sup>#</sup> compared with when PHL criteria were previously met

- If there is no significant change no action is required
- If there is a significant change follow the process described in <u>Follow-up</u> of this Appendix

<sup>#</sup>A 'significant' change in the subject's condition refers to a clinically relevant change in any of the individual liver biochemistry parameters (ALT, AST or total bilirubin) in isolation or in combination, or a clinically relevant change in associated symptoms. The determination of whether there has been a significant change will be at the discretion of the Investigator, this may be in consultation with the Protocol Officer if there is any uncertainty.

#### References

FDA Guidance for Industry (issued July 2009) 'Drug-induced liver injury: Premarketing clinical evaluation':

NCI Version Date: 05-06-2021 170(177) NSABP B-55/BIG 6-13

## **Appendix E** Acceptable Birth Control Methods

## Olaparib is regarded as a compound with medium/high foetal risk.

Women of childbearing potential who are sexually active, must agree with their partners, to the use of TWO highly effective forms of contraception in combination (as listed below). This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 1 month after the last dose of study drug, or they must totally/truly abstain from any form of sexual intercourse (see below). Please note that in breast cancer patients, hormonal contraception should only be used if considered appropriate by the investigator.

Male patients must use a condom during study treatment and for 3 months after the last dose of study drug when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Male patients should not donate sperm throughout the period of taking study treatment and for 3 months following the last dose of study drug.

## Acceptable non-hormonal birth control methods include

- Total/True abstinence: When the patient refrains from any form of sexual intercourse and this is in line with their usual and/or preferred lifestyle, this must continue for the total duration of the treatment period and for 1 month after the last dose of study drug for female patients, for 3 months after the last dose for male patients. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods, or declaration of abstinence solely for the duration of a trial) and withdrawal are not acceptable methods of contraception.]
- Vasectomised sexual partner plus male condom. With participant assurance that partner received post-vasectomy confirmation of azoospermia
- Tubal occlusion plus male condom
- IUD plus male condom. Provided coils are copper-banded

## Acceptable hormonal methods

- Etonogestrel implants (e.g., Implanon, Norplan) PLUS male condom
- Normal and low dose combined oral pills PLUS male condom
- Norelgestromin / EE transdermal system PLUS male condom
- Intravaginal device (e.g., EE and etonogestrel) PLUS male condom
- Cerazette (desogestrel) PLUS male condom. Cerazette is currently the only highly efficacious progesterone based pill.
- Hormonal shot or injection (e.g., Depo-Provera) PLUS male condom
- Intrauterine system [IUS] device (e.g., levonorgestrel releasing IUS Mirena®) PLUS male condom

NCI Version Date: 05-06-2021 171(177) NSABP B-55/BIG 6-13

## **Appendix F ECOG Performance Status**

## **Example of Performance Status (ECOG SCALE)**

| DESCRIPTION | ECOG GRADE |
|---|---|
| Fully active, able to carry on all pre-disease performance without restriction. | 0 |
| Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, i.e. light housework, office work. | 1 |
| Ambulatory and capable of self care, but unable to carry out any work activities. Up and about more than 50% of waking hours. | 2 |
| Capable of only limited self care, confined to bed or chair more than 50% of waking hours. | 3 |
| Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. | 4 |

NCI Version Date: 05-06-2021 172(177) NSABP B-55/BIG 6-13

# Appendix G Patient Reported Outcomes (FACIT-Fatigue, EORTC QLQ-C30)

## **FACIT Fatigue Scale (Version 4)**

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the <u>past 7 days</u>.

| | | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| НІ7 | I feel fatigued | . 0 | 1 | 2 | 3 | 4 |
| HI12 | I feel weak all over | . 0 | 1 | 2 | 3 | 4 |
| Anl | I feel listless ("washed out") | . 0 | 1 | 2 | 3 | 4 |
| An2 | I feel tired | . 0 | 1 | 2 | 3 | 4 |
| An3 | I have trouble starting things because I am tired | . 0 | 1 | 2 | 3 | 4 |
| An4 | I have trouble finishing things because I am tired | 0 | 1 | 2 | 3 | 4 |
| An5 | I have energy | 0 | 1 | 2 | 3 | 4 |
| An7 | I am able to do my usual activities | 0 | 1 | 2 | 3 | 4 |
| An8 | I need to sleep during the day | 0 | 1 | 2 | 3 | 4 |
| An12 | I am too tired to eat | 0 | 1 | 2 | 3 | 4 |
| An14 | I need help doing my usual activities | 0 | 1 | 2 | 3 | 4 |
| An15 | I am frustrated by being too tired to do the things I want | | | | | |
| | to do | 0 | 1 | 2 | 3 | 4 |
| An16 | I have to limit my social activity because I am tired | 0 | 1 | 2 | 3 | 4 |

English (Universal)
Copyright 1987, 1997
16 November 20
Page 1 o

NCI Version Date: 05-06-2021 173(177) NSABP B-55/BIG 6-13



## EORTC QLQ-C30 (version 3)

We are interested in some things about you and your health. Please answer all of the questions yourself by circling the number that best applies to you. There are no "right" or "wrong" answers. The information that you provide will remain strictly confidential.

| You | ase fill in your initials: or birthdate (Day, Month, Year): day's date (Day, Month, Year): 31 | | | | |
|---|---|---|---|---|---|
| | 10 | Not at | A<br>Little | Quite<br>a Bit | Very |
| I. | Do you have any trouble doing strenuous activities,<br>like carrying a heavy shopping bag or a suitcase? | 1 | 2 | 3 | 4 |
| 2. | Do you have any trouble taking a long walk? | 1 | 2 | 3 | 4 |
| 3. | Do you have any trouble taking a short walk outside of the house? | 1 | 2 | 3 | 4 |
| 4. | Do you need to stay in bed or a chair during the day? | 1 | 2 | 3 | 4 |
| 5. | Do you need help with eating, dressing, washing yourself or using the toilet? | 1 | 2 | 3 | 4 |
| Du | uring the past week: | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
| 6. | Were you limited in doing either your work or ther daily activities? | ) 1 | 2 | 3 | 4 |
| 7. | Were you limited in pursuing your hobbies or other leisure time activities? | 1 | 2 | 3 | 4 |
| 8. | Were you short of breath? | 1 | -2) | 3 | 4 |
| 9. | Have you had pain? | 1 | 1/2 | 3 | 4 |
| 10. | Did you need to rest? | | 2 | 1 | 4 |
| 11. | Have you had trouble sleeping? | 1 | 2 | 3 | 4 |
| 12. | Have you felt weak? | 1 | 2 | 3 | 4 |
| 13. | Have you lacked appetite? | 1 | 2 | 3 | 4 |
| 14. | Have you felt nauseated? | 1 | 2 | 3 | 4 |
| 15. | Have you vomited? | 1 | 2 | 3 | 4 |
| 16. | Have you been constipated? | 1 | 2 | 3 | 4 |

Please go on to the next page

NCI Version Date: 05-06-2021 174(177) NSABP B-55/BIG 6-13

| During the past week: | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|
| 17. Have you had diarrhea? | 11 | 2 | 3 | 4 |
| 18. Were you tired? | 1 | 2 | 3 | 4 |
| 19. Did pain interfere with your daily activities? | 1 | 2 | 3 | 4 |
| 20. Have you had difficulty in concentrating on things,<br>like reading a newspaper or watching television? | 1 | 2 | 3 | 4 |
| 21. Pid you/feel tense? | 1 | 2 | 3 | 4 |
| 22. Die you worry? | 1 | 2 | 3 | 4 |
| 23. Did you feel irritable? | 1 | 2 | 3 | 4 |
| 24. Did you feel depressed? | 1 | 2 | 3 | 4 |
| 25. Have you had difficulty remembering trings? | 1 | 2 | 3 | 4 |
| Has your physical condition or medical treatment interfered with your <u>family</u> life? | 1 | 2 | 3 | 4 |
| Has your physical condition or medical treatment interfered with your <u>social</u> activities? | 1 | 2 | 3 | 4 |
| 28. Has your physical condition or medical treatment caused you financial difficulties? | 1 | 2 | 3 | 4 |

# For the following questions please circle the number between 1 and 7 that best applies to you

| 29. | How | would | you r | rate you | r overall health | during the | past | week? |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

1 2 3 4 5

Very poor

30. How would you rate your overall quality of life during the past week?

1 2 3 4 5 6 7

Very poor Excellent

© Copyright 1995 EORTC Quality of Life Group. All rights reserved. Version 3.0



NCI Version Date: 05-06-2021 175(177) NSABP B-55/BIG 6-13

## **Appendix H** CPS & EG Score

Calculation instructions: Add the points for Clinical Stage + Pathologic Stage + ER status + Nuclear grade to derive a sum (CPS&EG score) between 0 and 6.

Table 18 Point assignments for the CPS + EG staging system

| Stage/feature | | Points |
|---|---|---|
| | I | 0 |
| | IIA | 0 |
| Clinical Stage | IIB | 1 |
| (AJCC staging <sup>1</sup> ) | IIIA | 1 |
| | IIIB | 2 |
| | IIIC | 2 |
| | 0 | 0 |
| | I | 0 |
| | IIA | 1 |
| Pathologic Stage (AJCC staging <sup>1</sup> ) | IIB | 1 |
| (AJCC staging) | IIIA | 1 |
| | IIIB | 1 |
| | IIIC | 2 |
| Receptor status | ER negative <sup>2</sup> | 1 |
| Nuclear grade <sup>3</sup> | Nuclear grade 3 | 1 |

AJCC: American Joint Committee on Cancer (<a href="https://cancerstaging.org/Pages/default.aspx">https://cancerstaging.org/Pages/default.aspx</a>)

<sup>&</sup>lt;sup>2</sup> ER: Estrogen receptor; definitions for ER negativity see eligibility criteria <u>section</u> <u>4.1.4.a</u>

In the unlikely situation nuclear grade cannot be determined, regular histologic grade should be used; if only Nottingham overall grade is reported, the Nottingham overall grade must be 9 to be scored as 1 point in the CPS&EG score (<a href="http://pathology.jhu.edu/breast/grade.php">http://pathology.jhu.edu/breast/grade.php</a>).







## Statistical Analysis Plan

Drug Substance Olaparib (AZD2281)

Study Code D081CC00006

Study Number BIG 6-13, NSABP B-55

Edition Number 3.0

Date

12<sup>th</sup> June 2019

A randomised, double-blind, parallel group, placebo-controlled multicentre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy

A randomised, double-blind, parallel group, placebo-controlled multicentre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy

AstraZeneca Study Statistician

A randomised, double-blind, parallel group, placebo-controlled multi-centre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy

AstraZeneca Global Product
Statistician

A randomised, double-blind, parallel group, placebo-controlled multicentre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy

| Frontier Science Statistician | |
|-------------------------------|-------------------------------|
| | Frontier Science Statistician |

A randomised, double-blind, parallel group, placebo-controlled multi-centre Phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA1/2* mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant chemotherapy

NRG Oncology Statistician

#### VERSION HISTORY

## Version 3.0 Final, [12th June 2019]

Substantial updates following protocol amendment (Protocol edition 5 dated 18 May 2018), discussions within the stats sub-team and AZ review of table shells.

The following sections are added or updated from SAP version 2.0:

- Section 1.3 and Section 5 Increase sample size to 1800 with 90% power and Table 4 Actual accrual pattern
- Section 1.4 Data cut-off interim analysis
- Section 2.1, 3.3.8 and 4.2.11 Pharmacokinetics (PK) analysis
- Section 2.1 Only patients with a signed informed consent will be included in the analysis sets
- Section 2.2 Important protocol deviations and 'deviation bias' sensitivity analysis.
- Section 2.2 Updated dispensing errors text, kit IDs are not available.
- Section 3.1 Censoring at 0.5 days for special cases, hierarchy of IDFS event categories and incidence of new cancers
- Section 3.3.1 Removed section on OAEs, OAEs have not been defined on Olympia as AZ do not have access to the data.
- Section 3.3.1- Adverse events section updated to match protocol version 5 (Section 6.4.3 Recording of adverse events).
- Section 3.3.1.1 Adverse events of special interest updated to match protocol version 5 (Section 6.4.3 Recording of adverse events).
- Section 3.3.2 and 3.3.3 Treatment exposure and dose intensity, due to eCRF design missed or forgotten doses within an individual day are not captured.
- Section 3.3.2 Included derivations for cumulative exposure over time, and exposure by dose.
- 4.2.1: Confidence intervals section included to describe what CI will be presented for each endpoint
- Section 4.2.2, 4.2.3 and 4.2.4 added.
- Section 4.2.5 Added table shell for fallopian tube history, time from diagnosis to randomisation and post-event treatments/radiotherapy/surgery.
- Section 4.2.3.1 Re-included AZ's preferred method for the pooling of the stratification factors.
- Section 4.2.7.2 Sensitivity analysis added: Incomplete follow-up, important protocol deviations, unadjusted analysis and interval censored Cox regression.
- Section 4.2.7.2 Interval censoring sensitivity analysis details of analysis method included.
- Section 4.2.7.2 Sensitivity analysis removed: Incomplete follow-up

- Section 4.2.7.3 CPS+EG score comes directly from the eCRF and data management check if the score is correct. Table 8 point assignments for the CPS+EG score derivation is obsolete and therefore deleted.
- Section 4.2.7.3 Expanded subgroup analyses methods.
- Section 4.2.7.3 pvalue for interaction to be assessed at 10% for purpose of hypothesis generation.
- Section 4.2.7.4 Added more detail on the global interactions
- Section 4.2.9 Expanded details on Fine and Gray models using SAS 9.4
- Section 4.2.10 Text on PRO consent included, included NRG updates to the PRO section
- Section 4.2.11 Specified LOQ is 0.0005 μg/mL
- Section 4.2.13 Summary of long term tolerability, analyses originally described for AESI are to be done for nausea, vomiting, anaemia, neutropenia, thrombocytopenia, and fatigue and asthenia
- Section 4.2.16 Central pathology result time point for analysis
- Section 4.2.13 Summary of AESI > 30days included
- Section 4.2.13 Updated the Hy's law section
- Section 4.2.13– Deaths section revised
- Section 4.2.14 Modifications replaced with interruptions and reductions
- Throughout Updated text for inadvertent randomisation to be clear that they had no follow-up nor treatment
- Section 4.2.9 Males excluded from analyses of new primaries that they are not at risk for.
- Section 6.1 Defence of censoring at 0.5 days.
- Appendix A Event prediction (survival model) for protocol amendment (protocol version 5.)
- Appendix D Contains the GailSimon macro
- Appendix E Included text on central pathology results
- Changed b.i.d to be bd throughout in line with AZ Olaparib studies
- References added for GailSimon macro, R packages for non-proportional hazards and for Greenwoods formula.
#### OlympiA SAP – Summary of Changes from V1 to V2

In line with the protocol edition 2 the number of subjects was increased, the resulted in updates to the following sections;

- 1.3 Number of subjects,
- Table 4 Estimated Accrual Pattern
- Added Table 5 Estimated Annual Hazard Rates
- Added Section on Revised Accrual Pattern with Tables 10-20
- 1.2 Study design
- 4.2.3.1 Primary analysis
- 4.2.6.3 Sample size consideration for PRO endpoints
- 5. Interim analysis
- Added Section 8 Appendix A

Other changes not relating to the increase in sample size include;

- 2.1 Added Definition of PK dataset
- 3.1.4 Added incidence of new primary fallopian tube cancer and new primary peritoneal cancer
- 4.2.1 Added section on Demographics and baseline characteristic data (moved from previous 4.2.8)

Under 4.2.3 Primary Endpoint Invasive Disease Free Survival IDFS, added headers to existing text for:

- 4.2.3.2 Sensitivity Analyses
- 4.2.3.3 Subgroup Analyses
- 4.2.3.4 Analysis of Interactions
- 4.2.5 Added Contralateral Invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, primary fallopian tube cancer and new primary peritoneal cancer
- 4.2.7 Added Pharmacokinetic Analysis
- 4.2.12 Added Imputation for missing/ partial dates

Added Section 9 Appendix B

Added Section 10 Appendix C

## **TABLE OF CONTENTS**

### **PAGE**

| | TITLE PAGE | 1 |
|---|---|---|
| | SIGNATURE OF STUDY STATISTICIAN | 2 |
| | SIGNATURE OF GLOBAL PRODUCT STATISTICIAN | 3 |
| | SIGNATURE OF GLOBAL PRODUCT STATISTICIAN | 4 |
| | SIGNATURE OF GLOBAL PRODUCT STATISTICIAN | 5 |
| | TABLE OF CONTENTS | 8 |
| 1. | STUDY DETAILS | 15 |
| 1.1 | Study Objectives | 15 |
| 1.2 | Study Design | 16 |
| 1.3 | Number of subjects | 29 |
| 1.4 | DCO Interim analysis | 30 |
| 2. | ANALYSIS SETS | 30 |
| 2.1 | Definition of analysis sets Full Analysis Set Safety Analysis Set PRO analysis set PK analysis set | 30<br>31 |
| 2.2 | Violations and deviations | 32 |
| 3. | PRIMARY AND SECONDARY VARIABLES | 34 |
| 3.1<br>3.1.1<br>3.1.2<br>3.1.3<br>3.1.4 | Outcome variables Invasive Disease Free Survival Overall Survival Distant disease free survival (DDFS). Incidence of contralateral invasive breast cancer, contralateral non- | 34 |
| 3.1.4 | invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer | 38 |
| 3.2<br>3.2.1<br>3.2.2 | Patient reported outcome variables FACIT-Fatigue EORTC QLQ-C30 | 39 |
| 3.3<br>3.3.1<br>3.3.1.1 | Safety | 40 |

| Study Code E<br>Study Numbe<br>Edition Numb | | |
|---|---|---|
| Date 27 May 3.3.2 | Treatment exposure | 42 |
| 3.3.3 | Dose intensity | |
| 3.3.4 | Laboratory data | |
| 3.3.5 | ECGs | |
| 3.3.6 | Vital signs | |
| 3.3.7 | General consideration for safety assessments | |
| 3.3.8 | PK variables | |
| 3.4 | Resource use | 47 |
| 4. | ANALYSIS METHODS | 47 |
| 4.1 | General principles | 48 |
| 4.2 | Analysis methods | 48 |
| 4.2.1 | Confidence intervals at the interim analysis | |
| 4.2.2 | Median clinical follow-up | |
| 4.2.3 | Kaplan-Meier estimates of IDFS | |
| 4.2.4 | Percentages of invasive disease free subjects at yearly intervals | |
| 4.2.5 | Demographic and baseline characteristics data | |
| 4.2.6 | Multiplicity | |
| 4.2.7 | Primary endpoint - Invasive Disease-Free Survival (IDFS) | |
| 4.2.7.1 | Primary Analysis | |
| 4.2.7.2 | Sensitivity Analyses for IDFS | 55 |
| 4.2.7.3 | Subgroup analyses | |
| 4.2.7.4 | Analysis of interactions | |
| 4.2.8 | Overall survival (OS) and Distant disease free survival (DDFS) | |
| 4.2.9 | Contralateral invasive breast cancer, contralateral non-invasive breast | |
| | cancer, new primary ovarian cancer, primary fallopian tube cancer and | |
| | new primary peritoneal cancer | |
| 4.2.10 | Analysis of patient reported outcomes | |
| 4.2.10.1 | Hypotheses and objectives | |
| | Administration of patient-completed questionnaire | |
| 4.2.10.3 | Statistical considerations for patient reported outcomes | |
| 4.2.11 | Pharmacokinetic analysis | |
| 4.2.11.1 | PK level deviations | |
| 4.2.12 | Exploratory analyses | |
| 4.2.13 | Safety | |
| 4.2.14 | Treatment exposure | |
| 4.2.15 | Imputation for Missing/Partial Dates | |
| 4.2.16 | Central pathology result timepoint for analysis | 80 |
| 5. | INTERIM ANALYSES | 80 |
| 6. | CHANGES OF ANALYSIS FROM PROTOCOL | 84 |
| 6.1 | Censoring of patients not at risk for disease evaluated | 84 |
| 7. | REFERENCES | 86 |

Statistical Analysis Plan

Drug Substance Olaparib (AZD2281) Study Code D081CC00006 Study Number BIG 6-13, NSABP B-55 Edition Number 3.0 Date 27 May 2019 APPENDIX A......89 8. 9. APPENDIX B......90 10. APPENDIX C 91 APPENDIX D......92 11. 12. APPENDIX E 94 12.1 12.2 Derivation of Central pathology results from the data provided by IEO......94 12.3 12.3.1 Considerations 95 12.3.2 Identifying the central pathology result ......96 LIST OF TABLES Study Schedule - Screening (PART 1 and PART 2) ......20 Table 1 Table 2 Table 3 Table 4 Table 5 Summary of Outcome Variables and Analysis Populations......31 Table 6 Table 7 Formal Statistical Analyses to be Conducted 50 Table 8 Table 9 Table 10 Summary of 2-sided significance levels and total alpha spend Table 11 Example of patient who permanently discontinued during a dose interruption, documented on eCRF page "Administration of Olaparib/Placebo"......90 Table 12 IEO data HR status (ER & PgR) and HER2 results (See DTS) ................94 Table 13 Derivations for classifications of HR status and HER2 results for

Statistical Analysis Plan

## **LIST OF FIGURES**

| Figure 1 | Study Flow Chart | 19 |
|----------|--------------------------------------------------------|----|
| Figure 2 | Screening Plan | 20 |
| Figure 3 | Multiple Testing Procedure | 53 |
| Figure 4 | Examples of dose intensity for olaparib/placebo dosing | 91 |

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

The following abbreviations and special terms are used in this study Statistical Analysis Plan.

| Abbreviation or special term | Explanation |
|---|---|
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AML | Acute Myeloid Leukaemia |
| AST | Aspartate aminotransferase |
| bd. | Twice daily |
| BIG | Breast International Group |
| BP | Blood pressure |
| BRCA | Breast cancer susceptibility gene |
| CI | Confidence Interval |
| CNS | Central nervous system |
| CPS+EG | Clinical stage (CS), estrogen receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS)- a disease scoring system |
| CRF (eCRF) | Case Report Form (electronic/paper) |
| CSP | Clinical Study Protocol |
| CSR | Clinical Study Report |
| CT | Computerised Tomography |
| CTCAE | Common Terminology Criteria for Adverse Event |
| CTEP | Cancer Therapy Evaluation Program |
| DBP | Diastolic blood pressure |
| DCO | Data cut off |
| DDFS | Distant Disease-Free Survival |
| DNA | Deoxyribonucleic acid |
| ECG | Electrocardiogram |
| ECOG performance status | Eastern Cooperative Oncology Group: a performance status using scales and criteria to assess how a patient's disease is progressing |
| eCRF | Electronic case report form |

| Abbreviation or special term | Explanation |
|---|---|
| EORTC QLQ-C30 | The European Organisation for Research and Treatment of Cancer -Quality of Life Questionnaire-Core questions 30 |
| ER | Estrogen receptor |
| FACIT-Fatigue | Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue<br>Measurement System |
| FAS | Full Analysis Set |
| FFPE | Formalin Fixed Paraffin Embedded |
| FDA | Food and Drug Administration |
| gBRCA mutation or gBRCAm | The term "gBRCA mutation" is used to refer to a germline BRCA1 or BRCA2 mutation classified as "deleterious" or "suspected deleterious" in accordance with the American College of Medical Genetics and Genomics recommendations for standards for interpretation and reporting of sequence variants |
| GCP | Good clinical practice |
| HER2 | Human Epidermal Growth Factor Receptor 2 |
| HR | Hazard Ratio |
| HRQoL | Health Related Quality of Life |
| ID | Identifier |
| IDFS | Invasive Disease-Free Survival |
| IDMC | Independent Data Monitoring Committee |
| IIBTR | Ipsilateral invasive breast tumour recurrence |
| IPD | Important protocol deviation |
| IQR | Inter-quartile range |
| ITT | Intention To Treat |
| IVRS | Interactive Voice Response System |
| IWRS | Interactive Web Response System |
| KM | Kaplan-Meier |
| MDS | Myelodysplastic Syndrome |
| MMRM | Mixed Model for Repeated Measures |
| MRI | Magnetic Resonance Image |
| MTP | Multiple Testing Procedure |
| NSABP | National Surgical Adjuvant Breast and Bowel Project |

| Abbreviation or special term | Explanation |
|---|---|
| NONMEM | NON-linear Mixed Effects Modelling |
| OS | Overall Survival |
| PARP | Polyadenosine 5'diphosphoribase [poly (ADP ribose)] polymerisation |
| pCR | Pathologic Complete Response |
| PGx | Pharmacogenetic research |
| PMG | Precision Medicin and Genomics |
| PID | Percentage Intended Dose |
| PK | Pharmacokinetics |
| PRO | Patient Reported Outcome |
| PgR | Progesterone receptor |
| QOL | Quality of Life |
| RDI | Relative Dose Intensity |
| REML | Restricted Maximum Likelihood |
| RPSFT | Rank Preserving Structural Failure Time |
| SAE | Serious adverse event (see definition in CSP Section 6.4.2). |
| SBP | Systolic blood pressure |
| SD | Standard Deviation |
| STEEP | Standardised Terms for Efficacy Endpoints |
| Study treatment | Study treatment is the treatment to which patient was randomised. In this study it is either olaparib or placebo |
| TNBC | Triple negative breast cancer |
| ULN | Upper Limit of Normal |

#### 1. STUDY DETAILS

### 1.1 Study Objectives

#### **Primary:**

The primary objective is to assess the effect of adjuvant treatment with olaparib on Invasive Disease Free Survival (IDFS).

#### **Secondary:**

The secondary objectives of this study are:

- 1 To assess the effect of adjuvant treatment with olaparib on Overall Survival (OS).
- 2 To assess the effect of adjuvant treatment with olaparib on Distant Disease Free Survival (DDFS).
- To assess the effect of adjuvant treatment with olaparib on the incidence of new primary contralateral breast cancers (invasive and non-invasive), new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer.
- To assess the effect of olaparib on the patient reported outcomes using the FACIT-Fatigue and EORTC QLQ-C30 questionnaires.
- To assess the efficacy of olaparib in patients identified as having a deleterious or suspected deleterious variant in either of the *BRCA* genes using variants identified with current and future germline *BRCA* mutation assays (gene sequencing and large rearrangement analysis).
- 6 To determine the exposure to olaparib (in plasma) in patients receiving olaparib as adjuvant therapy as part of the PK analysis.

#### Safety:

To assess the safety and tolerability of adjuvant treatment with olaparib





## 1.2 Study Design

This is a randomised, double-blind placebo controlled multi-centre, phase III study to assess the efficacy and safety of olaparib versus placebo as adjuvant treatment in patients with germline *BRCA*1/2 mutations and high risk HER2 negative primary breast cancer who have completed definitive local treatment and neoadjuvant or adjuvant treatment.

Patients will be randomised in a 1:1 ratio to either olaparib or placebo. Randomisation will use permuted blocks and will be stratified by hormone receptor status (ER and/or PgR

positive/HER2 negative versus TNBC), by prior neoadjuvant versus adjuvant chemotherapy, and prior platinum use for breast cancer (yes versus no).

Patients will be randomised to one of the following treatments:

- 12 months treatment with olaparib tablets p.o. 300 mg twice-daily (two 150 mg tablets in the morning and two 150 mg tablets in the evening)
- 12 months treatment with matching placebo tablets p.o. twice daily (two tablets in the morning and two tablets in the evening)

Randomised patients will receive study treatment for up to a maximum of 12 months. All patients will have safety assessments every 2 weeks during the first month, every 4 weeks for the following 5 months (up to week 24) and 3 monthly for the remaining 6 months of study treatment, plus 30 days after its discontinuation.

All randomised patients will have clinical assessment visits for approximately 10 years following their randomisation into the study, or until an IDFS endpoint due to a breast cancer related distant relapse, whichever comes first. Efficacy assessments (medical history and physical examination) will be performed on a 3 monthly basis during the first 2 years following end of study treatment, followed by 6 monthly assessments for years 3, 4 and 5 and annually thereafter. All patients will have a mammogram and/or breast MRI annually for approximately 10 years beginning 6 months (24 weeks) after day 1. They then enter the survival follow-up phase of the trial, which will continue until 10 years after the last patient is randomised. No clinic visits will be required during the survival follow-up phase; information may be collected via telephone, medical records and death registries.

This is a collaborative study being coordinated worldwide by the Breast International Group (BIG) in partnership with Frontier Science (FS), NRG Oncology (NCI supported National Clinical Trials Network Group), AstraZeneca (AZ) and Merck & Co (Merck). Two versions of the protocol have been written to cover this global adjuvant breast cancer study. One protocol version covers all patients recruited outside of the US (where AZ is the sponsor) and one protocol version covers patients recruited within the US (where NRG Oncology is the sponsor). The two versions of the protocol are identical in terms of study objectives and scientific content and only differ in logistical content appropriate for the country(ies) they cover (i.e. drug distribution, mechanisms for SAE reporting during the study, etc.). It is expected that approximately 230 patients will be randomised under the US protocol and approximately 1570 patients will be randomised under the non-US protocol.

The study will be conducted in approximately 25 countries worldwide. Approximately 700 centres (in the US and rest of the world countries) will be initiated to randomise the total 1800 patients. Additional countries and sites may be added dependent on recruitment rates.

The trial will use one randomisation system and report as one single study. The initial collection of the patients' data will be done using two databases (one for the US patients and one for all other patients outside of the US). The two databases will be set up using the same

standards and eCRFs to ensure consistency in the data collection. The data from both databases will be combined into a single consolidated database at regular, pre-specified intervals. All study endpoints as well as reports for periodic review by the Independent Data Monitoring Committee (IDMC) will be analysed and reported from the single combined reporting database, held by Frontier Science on behalf of BIG.

Approximately, 150 randomised patients will be analysed for pharmacokinetic (PK) at those sites that have confirmed that they are able to collect the PK assessment samples. PK sampling will be performed in a subset of patients who sign an optional PK Informed consent.

The study flow chart is shown in Figure 1 and the screening plan in Figure 2. Screening schedules are detailed in Table 1 and the study schedule is detailed in Table 2 and Table 3 below.

#### Figure 1 Study Flow Chart

ICF for patients with unknown *BRCA* status to undergo central *BRCA* testing during, or prior to, neoadjuvant/adjuvant chemotherapy



Figure 2

**Screening Plan** 

#### Screening PART 1- Patients with Unknown gBRCA Mutation Status:

• Only those patients who **do not** know their gBRCA mutation status prior to entry in to the study

These patients will undergo screening assessments as described for PART 1 in Table 1. Screening PART 1 is conducted to determine if the patient is considered **eligible to undergo the** *BRCA* **status blood test**. Once PART 1 has been successfully completed and patients have had a *BRCA* test, these patients will continue to PART 2 and have all procedures performed as described for PART 2 (see Table 1)

#### <u>Screening – PART 2 – ALL Patients (Patients with Known gBRCA Mutation Status)</u>:

- Those patients who already know their gBRCA mutation status **and** have a deleterious or suspected deleterious mutation to undergo screening assessments as described for PART 2 (see Table 1)
- Those patients originally with unknown gBRCA status who have completed screening PART 1 and now have a confirmed deleterious or suspected deleterious mutation should undergo screening assessments as described for PART 2 (see Table 1)

Table 1 Study Schedule - Screening (PART 1 and PART 2)

| Day | Any time prior, during or after neoadjuvant/adjuvant chemotherapy or radiotherapy PART 1 a (ONLY Patients requiring a gBRCA status Myriad test before randomisation) | -28 to 0 days PART 2 (Patients with confirmed gBRCA status by or if BRCA status is known prior to study entry j) |
|---|---|---|
| Informed consent | X bc | X <sup>j</sup> |
| Demographics (date of birth) | X | X |
| Medical and surgical history <sup>d</sup> | | X |
| Prior cancer therapies including radiotherapy | | X |
| Inclusion/exclusion criteria | X (all ** criteria) | X |
| ECOG Performance Status | | X |
| Physical examination | | X |
| Vital signs | | X |
| ECG <sup>f</sup> | | X <sup>g</sup> |

Table 1

### **Study Schedule - Screening (PART 1 and PART 2)**

| Day | Any time prior, during or after neoadjuvant/adjuvant chemotherapy or radiotherapy PART 1 a (ONLY Patients requiring a gBRCA status test before randomisation) | -28 to 0 days PART 2 (Patients with confirmed gBRCA status by or if BRCA status is known prior to study entry j) |
|---|---|---|
| Haematology / clinical chemistry/Coagulation ° | | X |
| Urinalysis <sup>h</sup> | | X |
| Pregnancy test i | | X |
| EORTC QLQ-C30 <sup>n</sup> | | X |
| FACIT-Fatigue <sup>n</sup> | | X |
| Blood sample for determination of <i>BRCA</i> status via | X | X e |
| Blood sample for assessment of current and future <i>BRCA</i> mutation assay(s) <sup>c</sup> | X | X e |
| Concomitant medications | | X |
| Archival tumour sample (FFPE) (mandatory if available) k | | X |
| Surgical tumour sample (FFPE) (post neoadjuvant chemotherapy (mandatory)) k | | X |
| Radiological assessment to exclude metastatic breast cancer (where applicable) <sup>1</sup> | | X |
| Family history of cancer | | X |
| Serious Adverse Events <sup>m</sup> | X (only SAEs due to study procedures) | X (SAEs only) |

| a | The time period is to allow those patients that require a | gBRCA sample to have the test taken and |
|---|---|---|
| | the results returned prior to randomisation | • |

b It is recommended that patients that require the *BRCA* sample testing are to be consented for *BRCA* testing and participation in the trial prior or during neoadjuvant/adjuvant chemotherapy prior to entering the study.

c Any patient who consents to study related gBRCA status testing, must also have a blood sample taken at the same time for the purpose of developing and validating a future mutation assay.

d Include history of blood transfusion within previous 120 days from start of study treatment and the reasons e.g. bleeding. Additionally CPS+EG score components should be collected (Clinical stage (CS), estrogen

- receptor status (E), nuclear grade (G), and post-treatment pathologic stage (PS)) for the non-pCR patients who received prior neoadjuvant chemotherapy. Instructions on how to calculate the CPS+EG score (Mittendorf et al 2011; Jeruss et al 2008) are provided in Appendix J of protocol edition 2.
- e Samples to be taken in screening PART 2 only for patients with known gBRCA mutation who have not completed PART 1.
- f ECG recordings should be performed once the patient has been in the supine position for at least 5 minutes.
- g ECG assessments to be completed within 28 days before randomisation.
- h Urinalysis (dipstick) should be performed at screening. After screening, urinalysis will only be required if clinically indicated.
- i Women who are not postmenopausal or have not undergone hysterectomy must have a negative urine or serum pregnancy test within 28 days prior to randomisation and a confirmatory test on Day 1 before starting study treatment. In the event of suspected pregnancy during the study, the test should be repeated and, if positive, the patient discontinued from study treatment immediately.
- j Patients for whom their gBRCA status is already known, should be consented to the study within 28 days prior to randomisation.
- k Mandatory for all randomised patients, i.e. for adjuvant patients this refers to the surgical specimen; for neoadjuvant patients, both the pre-treatment core biopsy and the surgical specimen with residual disease are requested but only one is mandatory. If the surgery tumour blocks are available, but cannot be submitted, sites may submit a portion of invasive tumour from the original block, either by taking at least one core of at least 3mm in diameter, or by splitting the original block in two parts, and re-embedding one in a new block for central submission. If blocks containing pre-neoadjuvant treatment core biopsies are available but cannot be submitted, sections mounted on glass slides prepared from the block can be provided. If tumour sample can't be provided as requested above or if it's not available, approval by Study Team for patient's entry into the trial is required. Sample will only be sent to the study bio-repository once the patient has been randomised.
- Patients considered at high risk of having disseminated disease (i.e. those with locally advanced disease, clinical N2-3 or pathological N1-3 with the exception of pN1a in adjuvant patients are expected to have a CT/MRI scan of the Thorax/Abdomen/Pelvis or any other area as clinically indicated and a bone scan at any point between diagnosis of the current breast cancer and randomisation to rule out metastatic breast cancer. (Note: PET/CT scan may be used as an alternative imaging technique and precludes the need for bone scan). If a patient does not have a mammogram or breast MRI within 12 months prior to screening part 1, then this assessment must be repeated prior to randomisation. Breast imaging should be performed on any remaining breast tissue.
  - To rule out metastatic breast cancer, patients with screening ALT/AST or ALP above institutional upper limit of normal should have liver ultrasound, CT or MRI at any time point between diagnosis of current breast cancer and randomisation. Screening bone scan is required if ALP and/or corrected calcium level are above the institutional upper limit. (Note: PET/CT scan may be used as an alternative imaging technique).
- m Serious adverse events must be captured from time of consent. In Screening PART 1 of the study only SAEs related to study procedure will be collected. In Screening PART 2 all SAEs will be collected.
- n EORTC OLO-C30 + FACIT-Fatigue will be collected prior to randomisation once eligibility is confirmed.
- o Coagulation analysis only required at baseline.

Study Schedule - On treatment (Year 1)

| Visit Number | 7 | m | 4 | 5-9<br>(Every 4<br>weeks) | 10-11<br>(Every 3 months<br>(14 weeks)) | Premature study treatment discontinuation § | Follow-up 30 days<br>after last dose of<br>study medication (all<br>patients) |
|---|---|---|---|---|---|---|---|
| Week | 0 | 2 | 4 | 8, 12, 16, 20, 24 | 38, 52 | | |
| Day | 1 | 15 | 29 | | | | |
| Visit Window | | <b>∓3</b> d | ±3d | ±1 week | ±2 week | +2 week | +2 week |
| Serum or urine pregnancy<br>test for women of<br>childbearing potential prior<br>to 1st dose of study<br>treatment | X a | | X | X | X | | X |
| ECOG performance status | q X | | | | | | |
| Vital signs | X b | | × | X (weeks 12 and 24 only) | X | X | X |
| Haematology / clinical chemistry c | X b,c | × | × | X | X | X | X |
| Recurrent/new cancers assessment (includes physical exam <sup>d</sup> , clinical signs and symptoms) | × | | | X (weeks 12 and 24 only) | × | × | X |
| Mammogram and/or breast<br>MRI (MRI preferred for<br>patients younger than 50<br>yrs) <sup>e</sup> | | | | X (week 24 only) | | | |
| Adverse Events | × | × | × | X | X | X | X |

Study Schedule – On treatment (Year 1)

| Visit Number | 2 | 3 | 4 | 5-9<br>(Every 4<br>weeks) | 10-11<br>(Every 3 months<br>(14 weeks)) | Premature study treatment discontinuation <sup>g</sup> | Follow-up 30 days<br>after last dose of<br>study medication (all<br>patients) |
|---|---|---|---|---|---|---|---|
| Week | 0 | 2 | 4 | 8, 12, 16, 20, 24 | 38, 52 | | |
| Day | 1 | 15 | 59 | | | | |
| Visit Window | | ±3d | ±3d | ±1 week | ±2 week | +2 week | +2 week |
| Concomitant medications including blood transfusions | × | × | X | X | X | X | X |
| Demographics <sup>j</sup> | X | | | | | | |
| EORTC QLQ-C30 | | | | X (week 24 only) | X (week 52 only) | | |
| FACIT-Fatigue | | | | X (week 24 only) | X (week 52 only) | | |
| Biomarker Blood 2 samples (mandatory) | Xi | | | | | | X |
| PGx Blood sample (optional) | X | | | | | | |
| Blood sample for PK<br>analysis (optional; after<br>signing PK Informed<br>consent) (subset of<br>patients) h | | | X | | | | |
| Blood biomarker samples<br>at disease recurrence<br>(Mandatory) | × | × | × | × | X | X | X |

Study Schedule – On treatment (Year 1)

| Visit Number | 2 | e | 4 | 5-9<br>(Every 4<br>weeks) | 10-11<br>(Every 3 months<br>(14 weeks)) | Premature study treatment discontinuation § | Follow-up 30 days<br>after last dose of<br>study medication (all<br>patients) |
|---|---|---|---|---|---|---|---|
| Week | 0 | 2 | 4 | 8, 12, 16, 20, 24 38, 52 | 38, 52 | | |
| Day | 1 | 15 | 29 | | | | |
| Visit Window | | <b>p</b> €∓ | р€∓ | ±1 week | ±2 week | +2 week | +2 week |
| Tumour sample at disease recurrence (Optional) k | X | X | X | X | X | X | X |
| Olaparib<br>dispensed/returned <sup>f</sup> | X | | × | X | X | X | |

Women who are not postmenopausal or have not undergone hysterectomy must have a negative urine or serum pregnancy test prior to first dose of study

f assessed within 7 days before randomisation, it does not need to be repeated on Day 1 of study treatment unless investigator believes that it is likely to have changed significantly.

Safety blood samples do not need to be repeated on Day 1 of study treatment if they have been assessed within 7 days before randomisation and which significantly. Safety blood samples are to be collected every 2 weeks during the first 4 weeks, then every 4 weeks until week 24 and then at weeks 38 must have been done at least 3 weeks after the last dose of chemotherapy, unless the investigator believes that they are likely to have changed and 52 of study treatment.

reatment is discontinued (data is not required to be captured on an eCRF, however any significant changes from baseline must be reported as an AE). Physical examination both local and general should be performed at day 1 and then at weeks 12, 24 and 38 and 52 post randomisation until study

Mammogram and/or breast MRI (MRI is preferred for patients younger than 50 years) to be performed at week 24 (6 months). Breast imaging should be performed on any remaining breast tissue.

Sufficient study treatment should be dispensed for at least each treatment period plus overage, however additional treatment can be dispensed to patients to last longer in accordance with local practice.

ba

followed by the 30 day follow-up visit and site staff completes relevant CRF pages as required. In case of premature treatment discontinuation only the visits where efficacy assessments are scheduled should be performed i.e. week 12, 24, 38, 52 (as applicable) in Year 1 and all visits in Year 2 onwards. herapies should be collected and recorded in the clinical database until IDFS endpoint is met due to breast cancer related distant relapse. The date of f a patient discontinues prior to completing 52 weeks of study treatment, the patient should have the study treatment discontinuation visit performed Collection of vital signs, AEs, haematology/clinical chemistry results and concomitant medications is no longer required. Information on endocrine liscontinuation, the reasons, and details of the following specific cancer therapies (first line treatment for first breast cancer recurrence and any

subsequent regimens containing PARP inhibitors or platinum received by the patient at any time) should also be recorded on the eCRF. In case the IDFS distant relapse and until 10 years after the last patient is randomised. In the IDFS endpoint is met due to other events, the patient will continue the study regimens containing PARP inhibitors or platinum received by the patient at any time), sites of metastases and any other new cancers. If a recurrent/new first. They will then enter the survival follow-up phase of the trial. During the annual survival follow-up phase, in addition to vital status, the following schedule until a breast cancer related distant relapse occurs or approximately 10 years following their randomisation into the study, whichever occurs endpoint is met due to breast cancer related distant relapse, the patient enters the survival follow-up phase and is assessed annually from the date of information will be collected (if available): specific cancer therapies (only first line treatment for first breast cancer recurrence and any subsequent cancer assessment is scheduled within 4 weeks of the study treatment discontinuation visit it can be performed at the 30-day follow-up visit.

PK sampling (optional) to be performed in a subset of patients. Sampling times: pre-dose (before morning dose) plus one sample in each of the following sampling windows: 0 to 0.5 h post dose, 0.5 to 1.5 h post dose, 3 to 6 h post dose and 6 to 12 h post dose (before evening dose) Blood samples (plasma and serum) for biomarker analysis should be collected on Day 1 prior to first dose of study treatment. Ч

The provision of tumour tissue is encouraged only if clinically appropriate and not considered detrimental to patient care and patient signed the Race and ethnicity data to be collected unless not allowed by local regulations. appropriate consent form.

Study Schedule - Follow-up Visits (Year 2 onwards)

Table 3

| Visit Number | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | Survival<br>Follow-up<br>(Every 12<br>months) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Year | | (4 | 2 | | 3 | | 4 | | 3 | | 9 | 7 | 8 | 6 | 10 | +11+ |
| Month | 15 | 18 | 21 | 24 | 30 | 36 | 42 | 48 | 54 | 09 | 99 | 78 | 06 | 102 | 114 | 126, 138,<br>etc. |
| Visit Window | | ±1month | onth | | | | ±2months | nths | | | | # | ±3months | ths | | ±3months |
| Recurrent/new cancers assessment (includes physical exam, clinical signs and symptoms) | X | × | × | × | × | × | × | X | × | × | × | × | × | × | X | |
| Mammogram and/or breast<br>MRI (MRI preferred for<br>patients younger than 50 yrs) <sup>a</sup> | | X | | | X | | × | | × | | × | X | X | × | X | |
| Subsequent cancer therapy <sup>b</sup> | X | X | X | X | X | × | × | × | X | X | X | X | X | X | X | pX |
| Overall survival assessment | | | | | | | | | | | | | | | | pX |
| EORTC QLQ-C30 | | × | | × | | | | | | | | | | | | |
| FACIT-Fatigue | | X | | X | | | | | | | | | | | | |
| Blood biomarker samples at disease recurrence (Mandatory) | X | X | X | × | × | X | X | X | × | × | × | × | × | × | X | |
| Tumour sample at disease recurrence (Optional) ° | X | × | X | X | X | × | × | × | X | × | × | X | X | X | X | |

| Visit Number | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 12 13 14 15 16 17 18 19 20 21 22 23 24 25 26 | Survival<br>Follow-up<br>(Every 12<br>months) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Year | | 7 | | | 3 | | 4 | | 3 | | 9 | 7 | 8 | 6 | 6 7 8 9 10 | 11+ |
| Month | 15 | 18 | 21 | 24 | 30 | 36 | 42 | 48 | 54 | 09 | 99 | 78 | 06 | 102 | 114 | 15 18 21 24 30 36 42 48 54 60 66 78 90 102 114 126,138, etc. |
| Visit Window | | ±1month | onth | | | | $\pm 2$ months | nths | | | | # | ±3months | ths | | ±3months |
| SAE | X | X | × | × | × | × | × | × | × | × | × | × | × | × | x x x x x x x x x x x x x x x x x x x | X |

- Mammogram and/or breast MRI (MRI is preferred for patients younger than 50 years) to be performed every 12 months after the 6 months (24 weeks) scan, unless indicated otherwise. Breast imaging should be performed on any remaining intact breast. B
  - First line treatment for first breast cancer recurrence and any subsequent regimens containing PARP inhibitors or platinum received by the patient at any time need to be recorded. Information on endocrine therapies should be collected and recorded in the clinical database until IDFS endpoint is met due to reast cancer related distant relapse.
- The provision of tumour tissue is encouraged only if clinically appropriate and not considered detrimental to patient care and patient signed the appropriate consent form.
- During the survival follow-up phase, information (where available) on further subsequent cancer therapies (see footnote b), sites of metastases and any other new cancers will be collected in addition to vital status.
- completed the post treatment follow-up period (30 days). If an investigator learns of any SAEs, including death, at any time after a patient has completed the 30 days post treatment follow-up period, and he/she considers there is a reasonable possibility that the event is causally related to the study treatment, of the seriousness criteria is met which then requires to be reported as an SAE, see section 6.4.2 of the protocol edition 2. Any of these type of serious or after the 30 day follow-up period should be reported as an SAE. Non-melanoma skin cancers need to be reported as a non-serious AE unless at least one assessment of causality or knowledge of the treatment arm. If a patient develops MDS/AML full diagnostic details and classification should be provided information on new AEs or SAEs occurring to study patients. This includes new AEs/SAEs in patients still being followed up for survival but who have he investigator should report it according to SAE reporting procedures for this study. Any cases of MDS/AML or new primary malignancies occurring non-serious events need to be reported to AstraZeneca Patient Safety according to SAE reporting procedures for this study, regardless of investigator's After study treatment completion (i.e. after any scheduled post treatment follow-up period has ended) there is no obligation to actively report e.g. bone marrow and cytogenetic analysis reports, see Sections 5.5.6.3 and 6.4.5.5 of protocol edition 2. A questionnaire will be sent to any nvestigators reporting MDS/AML or new primary malignancies as an aid to provide detailed information on the case.

Date 12th June 2019

#### 1.3 Number of subjects

The primary endpoint of the study is invasive disease free survival (IDFS) and patients will be randomised 1:1 to either olaparib 300 mg bd or matching placebo.

Approximately, 1800 patients will be randomised into the study. If the true hazard ratio (HR) for the comparison of olaparib versus placebo (in terms of IDFS) is 0.7, then with 330 events the analysis of IDFS will have 90% power to demonstrate a statistically significant difference, assuming a 2-sided 5% significance level.

The primary analysis will be triggered by 330 IDFS events (required for overall 90% power to detect a HR at 0.7). The critical HR value at the primary analysis is 0.805.

The actual accrual pattern between June 2014 and February 2018 is shown in Table 4. It is estimated that 1800 patients will be randomised by April/May 2019, hence the study will take approximately 5 years to complete recruitment. (Around 230 patients in US and approximately 1570 patients in the Rest of World (RoW) countries).

Table 4 Actual accrual between June 2014 and February 2018

| Interval since start of randomisation (months) | Number of patients randomised in interval * | Cumulative<br>number of<br>patients<br>randomised | Average number of patients randomised per month in interval |
|---|---|---|---|
| 0 - 6 | 21 | 21 | 3.5 |
| 6 - 12 | 94 | 115 | 15.7 |
| 12 - 18 | 174 | 289 | 29.0 |
| 18 - 24 | 180 | 469 | 33.0 |
| 24 - 30 | 229 | 698 | 38.2 |
| 30 - 36 | 249 | 947 | 41.5 |
| 36 - 42 | 234 | 1181 | 39.0 |
| 42 - 45* | 118 | 1299 | 39.3 |

<sup>\*</sup> Note: 3-month interval: Dec 2017 to Feb 2018 inclusive

The primary analysis population will include all patients randomised (ITT). Subgroup analyses based on prior chemotherapy (adjuvant or neoadjuvant), prior platinum therapy (yes or no), and hormone receptor status (ER and/or PgR positive/HER2 negative versus TNBC) will be conducted to check for consistency in the treatment effect, whereby this analysis is considered supportive of the primary analysis in the overall population. Stratification factor values according to eCRFs will be used to define subgroups for the subgroup analyses.

During the trial, the Steering Committee will monitor the recruited patient population and actual event rate whilst remaining blinded to treatment allocation. If the data indicates that the original sample size assumptions are incorrect, such that achieving the required number of events with the current number of patients is not feasible, then in consultation with the IDMC a decision may be made to increase recruitment of patients into the trial to achieve the required 330 events.

An interim analysis for superiority will be triggered once 165 IDFS events have been observed in the first 900 patients recruited (see Section 5 for details). It is estimated that this analysis will occur approximately 5.4 years after the first patient is randomised.

## 1.4 DCO Interim analysis

The data cut-off (DCO) for the interim analysis is defined as the date that the 165<sup>th</sup> event confirmed by clinical exams, from the first 900 randomised patients, is reported in the database. Due to the reporting lag, this date will be later than the date when the 165<sup>th</sup> event is observed and confirmed in the clinic.

A programmatic data-cut will be applied to the OlympiA clinical database prior to the Interim and Final Analyses as defined in OlympiA datacut specification.docx .

#### 2. ANALYSIS SETS

#### 2.1 Definition of analysis sets

Only patients that signed the main informed consent form will be analysed, the analysis sets are defined as follows:

#### **Full Analysis Set**

Intention to treat (ITT): The primary statistical analysis of the efficacy of olaparib will include all randomised patients and will compare the treatment groups based on randomised treatment, regardless of the treatment actually received. Patients who were randomised but did not subsequently go on to receive study treatment are included in the Full Analysis Set (FAS).

For the interim analysis (see Section 5) two efficacy populations will be defined:

- ITT population: This will include all randomised patients and will compare the treatment groups based on randomised treatment, regardless of the treatment actually received. Note: it is anticipated that all patients will be randomised by the time of the interim analysis.
- 2 Mature cohort ITT population: This will include the first 900 randomised patients only and will compare the treatment groups based on randomised treatment, regardless of the treatment actually received. This analysis will be regarded as supportive, to aid

interpretation of the result in the ITT population based on interim data. Statistical significance is not required for the mature cohort population.

#### Safety Analysis Set

All safety data will be summarised by actual treatment received. All patients who received at least one dose of randomised study treatment, olaparib or placebo, will be included in the Safety Analysis Set. If a patient receives at least one dose of olaparib he/she will be included in the olaparib arm for safety summaries (e.g. olaparib arm will include patients randomised to olaparib who receive at least one dose of olaparib or placebo patients who receive at least one dose of olaparib in error at any time). If a patient randomised to olaparib receives only placebo treatment then he/she will be summarised as part of the placebo arm.

#### PRO analysis set

This population will comprise patients who consent to participate in the PRO assessment portion of the study, who start treatment and who provide evaluable baseline FACIT-Fatigue or EORTC QLQ-C30 data, where evaluable means that at least one sub-scale baseline score can be determined. Baseline is defined as the last result on or before the first day of study drug. For patients who are randomised but not treated, baseline will not be derived and they will be excluded from the PRO analysis set. Two sub-populations will be analysed dependent on whether they have evaluable baseline for the questionnaire being analysed. The PRO analysis will be summarised by planned treatment group.

#### PK analysis set

Approximately 150 patients randomised to olaparib/placebo will provide pharmacokinetic (PK) samples at those sites that have confirmed that they are able to collect the PK assessment samples. Placebo samples will not be analysed unless specified. PK sampling will be performed in a subset of patients who sign an optional PK informed consent.

The PK analysis set will comprise of patients who signed the optional PK informed consent form, were randomised to the olaparib arm, received at least one dose of study treatment, had at least one PK sample collected and did not violate or deviate from the protocol in ways that would significantly affect the PK analyses. The population will be defined by the Study Team Physician, Pharmacokineticist and Statistician prior to any analyses being performed and whilst blinded to treatment allocation.

Table 5 Summary of Outcome Variables and Analysis Populations

| Outcome Variable | Analysis set |
|---|---|
| Efficacy data Interim | |
| IDFS | FAS (ITT), Mature cohort (ITT) |
| IDFS, OS, DDFS, incidence of contralateral breast cancer, | FAS (ITT) |
| new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer and symptom/HRQoL endpoints | |

Table 5

#### **Summary of Outcome Variables and Analysis Populations**

| Outcome Variable | Analysis set |
|---|---|
| Efficacy data Final | FAS (ITT) |
| IDFS, OS, DDFS, incidence of contralateral breast cancer, | |
| new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer and symptom/HRQoL endpoints | |
| Demography | FAS (ITT) |
| PRO data | PRO |
| Pharmacokinetics data | PK |
| Safety data | |
| Exposure | Safety |
| Adverse Events | Safety |
| Lab measurements | Safety |
| Vital Signs | Safety |

#### 2.2 Violations and deviations

The important protocol deviations will be listed and summarised by randomised treatment group for the FAS. None of the deviations will lead to any patients being excluded from any of the primary analysis sets described in Section 2.1.

A per-protocol analysis is not planned, however a 'deviation bias' sensitivity analysis will be performed if the following criteria are met. Patients with important protocol deviations (IPDs) that may affect the efficacy of the trial therapy (as listed below) will be excluded if >10% of the randomised patients:

- Did not have the intended disease or indication or
- Did not receive any randomised therapy

The trigger for a sensitivity analysis will be determined following review of the protocol deviations ahead of database lock or data freeze for the interim analysis and final analysis. This will be documented prior to the analysis being conducted.

The following general categories will be considered as IPDs and be summarised and discussed in the CSR. Further detailed criteria are described in a separate Important Protocol Deviations Specification V6.0.

IPDs that may affect efficacy

- Not fulfilling criteria for high risk disease
- No histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast
- No documented germline mutation in BRCA1 or BRCA2
- Inadequate breast surgery and/or radiotherapy
- Inadequate axilla surgery
- Completed less than 6 cycles of neoadjuvant or adjuvant chemotherapy containing anthracyclines, taxanes or the combination of both
- Peri-operative chemotherapy, (patients who had both neoadjuvant and adjuvant therapy; 'unquantifiable risk of disease relapse')
- Evidence of metastatic disease (to include only those patients who had suspicion or confirmation of recurrence prior to randomisation)
- No staging or insufficient staging
- Prior PARP inhibitor use
- Prior cancer < 5 years ago including MDS/t-AML
- Randomized but did not receive any study treatment
- Received no study treatment whatsoever for a period of more than 7 days due to errors in dispensing of medication.
- Received an alternative study treatment to that which they were randomized
- Received prohibited concomitant medication
- Lack of confirmatory exams for events that count towards the analysis end points, efficacy and safety

#### <u>IPDs – GCP violations</u>

- GCP violation relating to informed consent
- GCP violation relating to serious adverse events
- GCP violation: other

The final classification will be made prior to database lock and all decisions will be made whilst blinded to study treatment allocation. For example, details of disallowed concomitant medication use will be reviewed by a physician using blinded data and may be determined as key.

Incorrect stratifications (i.e. patients for whom incorrect stratification information was provided at the time of randomisation) will be listed and summarised. In addition, any known treatment dispensing errors will also be listed and summarised. Dispensing errors, considered IPDs are described above.

Patients who receive the wrong treatment at any time will be included in the Safety Analysis Set as described in Section 2.1.

#### 3. PRIMARY AND SECONDARY VARIABLES

#### 3.1 Outcome variables

#### 3.1.1 Invasive Disease Free Survival

The primary endpoint of the trial is invasive disease free survival (IDFS), defined as the time from randomisation to date of first recurrence, where recurrence is defined as loco-regional, distant recurrence, new cancer or death from any cause. IDFS is further detailed according to the standardised terms for efficacy endpoints (STEEP) system definition (Hudis et al 2007) as one of the following:

- Ipsilateral invasive breast tumour recurrence (IIBTR): Invasive breast cancer involving the same breast parenchyma as the original primary.
- Regional invasive breast cancer recurrence: Invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast.
- Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or radiologically diagnosed as recurrent invasive breast cancer.
- Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
- Contralateral invasive breast cancer.
- Second primary non-breast invasive malignancies (i.e., excluding new in situ carcinomas of any site). Second primary non-breast invasive malignancies include hematologic malignancies and MDS. Squamous or basal cell skin cancers will not be counted as primary endpoint events.

Loco-regional recurrence of the disease (ipsilateral or regional invasive breast cancer) should be cytologically/histologically confirmed. Appropriate imaging (CT, MRI bone and/or PET scan) of the chest/abdomen/pelvis or any other area as clinically indicated should be performed at the time of local recurrence to exclude further spread of the disease. Distant recurrence should be diagnosed by radiological examination and/or histopathological confirmation when metastatic lesion is easily accessible for biopsy.

For confirmed local recurrence events, the earliest date of diagnosis based on an objective finding (physical exam, radiological/imaging assessment, and cytological/histopathological assessment) will be used to determine the time to event for the analysis but not the date of the first symptoms or blood analysis abnormality. For example, if a physical exam results in 'suspected' disease recurrence and disease recurrence is then confirmed by cytology/histology then the date of the physical exam will be used to derive the time to event.

For confirmed distant recurrence, the date of the earliest radiological/imaging examination or cytological/histopathological assessment linked to the diagnosis will be used to determine the time to event for the analysis (i.e. neither the symptoms or blood analysis, nor the physical exam, will be considered within the derivation of time to distant recurrence).

Invasive contralateral breast cancer or invasive non-breast secondary primary cancer should be confirmed by histopathological report. The date of the earliest objective finding related to diagnosis of the new cancer will be used as the date of new cancer for the analysis.

If multiple recurrence events are reported within 2 months of each other this is referred to as a simultaneous event and will be considered as a single event. In this situation, the worst case will be taken, as the event 'type' but the date of recurrence will be the earliest date of the multiple events. For example, if local and distant recurrence are reported within a 2-month period, then for the analysis and reporting of IDFS, the event type will be distant recurrence but the date of recurrence will be the earlier date of the two events.

If 2 recurrence events are reported but more than 2 months has elapsed between the events, then the events will be regarded as two separate recurrence events and the earlier event and corresponding date of event will be used in the derivation of IDFS (i.e. IDFS is based on the first recurrence event).

The hierarchy of event categories, from most to least severe (and with death without recurrence as last in hierarchy), will be as follows:

- CNS recurrences
- Distant visceral recurrence: lung, liver, pleural effusion
- Distant bone recurrence
- Other distant recurrence (assumed soft tissue)
- Regional recurrences
- Local recurrences
- Invasive contralateral breast cancer
- Second (non-breast) primary malignancy
- Death without recurrence
- If a patient dies during the study, and while being followed-up for efficacy, i.e. before the patient enters the survival follow-up only phase, and has no documented disease recurrence or invasive contralateral breast cancer or invasive non-breast secondary primary cancer then death will be regarded as an event and the date of death will be used to determine the patient's IDFS time.

Patients who have not had a recorded IDFS event at the time of the analysis will be censored at their last disease evaluation if efficacy follow-up is ongoing, or at the date of last contact if lost to follow-up, withdrawn from study or consent to survival follow-up only. For the purpose of the 10-year update, any patients completing the 10-year follow-up visit without recorded IDFS event will be censored at the 10-year follow-up visit. Disease evaluation includes mammogram and/or breast MRI (MRI preferred for patients younger than 50 years), other radiological/imaging examination or clinical examination (e.g. physical exam).

Patients will be censored at 0.5 days after randomisation under the following three circumstances:

- Patients who have had an event prior to randomisation.
- Patients who were identified as inadvertent randomisations (i.e. patient was randomised and the site noticed afterwards that they should not have been randomised, they have had no follow-up nor did they receive treatment).
- Patients who have withdrawn consent, received no treatment, and will not be providing any follow-up data.

#### 3.1.2 Overall Survival

Overall survival is defined as the time from the date of randomisation until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.

- Date of last contact given that the patient status is alive recorded within the survival follow-up module of the eCRF
- Date of randomisation
- Date of last contact
- NRG: "Date of last contact" on the "End of study" form
- RoW: "Date of last contact or death" on the "End of study" form
- Date of last disease evaluation
- Date of consent change for patients with "Partial withdrawal of consent, survival followup only"
- Date of withdrawal.

Patients will be censored at 0.5 days after randomisation under the following two circumstances:

- Patients who were identified as inadvertent randomisations (i.e. patient was randomised and the site noticed afterwards that they should not have been randomised, they have had no follow-up nor did they receive treatment).
- Patients who have withdrawn consent, received no treatment, and will not be providing any follow-up data.

#### 3.1.3 Distant disease free survival (DDFS)

DDFS will be defined as the time from randomisation until documented evidence of first distant recurrence of breast cancer or death from any cause. Distant recurrence will include the following events (as per STEEP system definition):

- Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or radiologically diagnosed as recurrent invasive breast cancer.
- Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
- Second primary non-breast invasive cancer.

Evidence of distant recurrence should be provided by either radiological examination or preferably by histopathological examination when metastasis is easily accessible for biopsy.

Second primary non-breast invasive cancer should be confirmed by histopathological report.

For the analysis of DDFS, the date of the confirmed DDFS event will use the earliest assessment date from the radiological and/or histological or cytological assessment. For example, if a patient has distant recurrence suspected by radiological examination which is later confirmed by biopsy, then the date of the radiological examination will be used as the date of event.

The hierarchy of event categories, from most to least severe (and with death without recurrence as last in hierarchy), will be as follows:

- CNS recurrences
- Distant visceral recurrence: lung, liver, pleural effusion
- Distant bone recurrence
- Other distant recurrence (assumed soft tissue)
- Second (non-breast) primary malignancy
- Death without recurrence

If multiple recurrence events are reported within 2 months of each other then this is referred to as a simultaneous event and will be considered as a single event. In this situation the worst case will be taken as the event 'type' but the date of recurrence will be the earliest date of the multiple events.

If 2 recurrence events are reported but more than 2 months has elapsed between the events, then the events will be regarded as two separate recurrence events and the earlier event and corresponding date of event will be used in the derivation of DDFS (i.e. DDFS is based on the first recurrence event).

Patients who do not have documented evidence of DDFS at the time of the analysis of DDFS will be censored at:

- Last disease evaluation if efficacy follow-up is ongoing
- Date of last contact if lost to follow-up, withdrawn from study or consent to survival follow-up only
- For the purpose of the 10 year update, any patient completing 10 year follow-up visit without recorded DDFS event will be censored at 10 year follow-up.

Disease evaluation includes mammogram and/or breast MRI (MRI preferred for patients younger than 50 years), other radiological/imaging examination or clinical examination (e.g. physical exam).

Patients will be censored at 0.5 days after randomisation under the following 3 circumstances:

- Patients who have had an event prior to randomisation, if the event was distant disease.
- Patients who were identified as inadvertent randomisations (i.e. patient was randomised and the site later realised that they should not have been randomised, they have had no follow-up nor did they receive treatment).
- Patients who have withdrawn consent, received no treatment, and will not be providing any follow-up data.

The first site of distant recurrence will be recorded and used in the analysis. Information on subsequent sites of recurrence will also be collected during follow up assessments to ensure as complete as possible information on distant recurrence is obtained.

# 3.1.4 Incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer

All patients should be followed for evidence of new primary breast cancers and all other cancers. This includes patients with a first event of local or distant recurrence as they might develop new cancers in the future. All new cancers will be collected for all patients not just the first new cancer.

Evidence of new contralateral breast cancer (invasive and non-invasive), and new ovarian, fallopian, or peritoneal cancers should be confirmed by clinical or radiological examination, with positive histology or cytology (confirmation of invasive tumour). The date of event will be taken as the earliest date from radiological, clinical and, histological or cytological exam (invasive disease only).

Time to new primary contralateral (invasive and non-invasive) breast cancer is defined as the interval between the date of randomisation and the date of the first occurrence of a new primary contralateral invasive breast cancer. Data analyses of new contralateral breast cancer (invasive and non-invasive) will exclude patients who have had bilateral mastectomy prior to randomisation.

Time to new ovarian cancers is defined as the interval between the date of randomisation and the date of the first occurrence of a new ovarian cancer, data analyses of new ovarian cancers will exclude patients who have had both ovaries removed prior to randomisation. Male patients will also be excluded from this analysis.

Time to new fallopian tube cancer is defined as the interval between the date of randomisation and the date of the first occurrence of a new fallopian tube cancer, data analyses of new fallopian tube cancers will exclude patients who have had both fallopian tubes removed prior to randomisation. Male patients will also be excluded from this analysis.

Time to new peritoneal cancer is defined as the interval between the date of randomisation and the date of the first occurrence of a new peritoneal cancer. Data analyses of new peritoneal cancer will include all patients in the ITT population with the exception of male patients, males will be excluded from this analysis.

Patients will be censored at 0.5 days after randomisation under the following 3 circumstances:

- Patients who have had an event prior to randomisation, if the event is the one being analysed.
- Patients who were identified as inadvertent randomisations (i.e. patient was randomised and the site later realised that they should not have been randomised, they have had no follow-up nor did they receive treatment).
- Patients who have withdrawn consent, received no treatment, and will not be providing any follow-up data.

#### 3.2 Patient reported outcome variables

Patient reported outcomes will be assessed based on the FACIT-Fatigue symptoms scale and the EORTC QLQ-C30 scale.

#### 3.2.1 FACIT-Fatigue

The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F Scale) is a 13-item questionnaire that assesses patient self-reported fatigue and its impact upon daily activities and function (Yellen et al 1997).

The FACIT-Fatigue scale is a validated instrument with a set method for scoring (FACIT-Fatigue Subscale Scoring Guidelines Version 4). The scale includes 13 items asking in different ways how the patients feels regarding being energetic, tired, weak or fatigue in the past 7 days with the patient selecting one of five categories of feeling levels ranging from "not at all" to "very much." Items #1 through #6 and items #9 through #13 are scored as follows: not at all=4; a little bit=3; somewhat=2; quite a bit=1; very much=0. Items #7 and #8 are reversed scored as follows: not at all=0; a little bit=1; somewhat=2; quite a bit=3; very much=4. The composite score is found by summing the scores for each of the 13 items. Thus, the composite score range is 0-52. The higher the score, the better the quality of life. A score of less than 30 indicates severe fatigue.

The FACIT-F scale was originally developed to evaluate fatigue associated with anaemia in cancer patients and has been used as an endpoint in clinical trials in various cancer populations including breast cancer and non-small cell lung cancer. Content validity of the FACIT-F has been demonstrated in a large sample of mixed cancer patients (n>300). Reliability (internal consistency, test-retest reliability, criterion validity, and responsiveness/sensitivity to change) of the FACIT-F have also been documented (Yellen et al 1997).

#### **3.2.2 EORTC QLQ-C30**

In this study patient-reported disease related symptoms and health-related quality of life (HRQoL) will be evaluated using the validated EORTC QLQ-C30 questionnaire (EORTC QLQ-C30 Scoring Manual 3<sup>rd</sup> edition). The EORTC QLQ-C30 questionnaire was developed to assess HRQoL and is the most commonly used cancer-specific tool in oncology. It has

undergone extensive testing and validation as well as detailed cross-cultural testing and validation and has been used in breast cancer trials.

The EORTC QLQ-C30 comprises 30 questions designed for all cancer types. Questions can be grouped into the following scales:

- 5 multi-item functional scales (physical, role, emotional, cognitive and social)
- 3 multi-item symptom scales (fatigue, pain, nausea vomiting)
- A 2-item global health status/QoL scale
- 5 single items assessing the following common cancer symptoms:
  - dyspnoea
  - loss of appetite
  - insomnia
  - constipation
  - diarrhoea
- 1 item on the financial impact of the disease.

All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high health/level of functioning, a high score for the global health status/QOL represents a high QOL, but a high score for a symptom scale /item represents a high level of symptomatology/problems.

The global health status/QOL score is based on two items (numbers 29 and 30) from the EORTC-QLQ-C30.

### 3.3 Safety

Safety and tolerability will be assessed for all randomised patients who received at least one dose of study treatment in terms of adverse events (AEs), serious adverse events (SAE), deaths, laboratory data and vital signs.

#### 3.3.1 Adverse events

Adverse events will be collected from time of signature of main informed consent\* throughout the treatment period up to and including the 30-day follow-up period. All ongoing and any new AEs/SAEs identified during the 30 calendar days follow up period after the last dose of study medication must be followed to resolution unless the event is considered by the

investigator to be unlikely to resolve, or the patient is lost to follow-up or in survival followup. Any medical condition (new or worsening of a pre-existing condition) that occurs post Screening PART 2 and is continuing at randomisation should be recorded in medical history in the eCRF as a medical condition current at randomisation. If the condition worsens post randomisation, this should be recorded as an AE/SAE in the eCRF with start date as the date the grade worsened and the new grade should be reported on the AE form. The AE/SAE would be considered to have resolved when it resolves to the baseline grade, not to zero. Any medical condition considered of clinical relevance (new or worsening of a pre-existing condition) that occurs post consent for PART 2 and resolves prior to randomisation should also be recorded as medical history. Any AE happening from randomisation to the 30-day follow-up period should be reported on the AE form in the eCRF. If an investigator learns of any SAEs, including death, at any time after a patient has completed 30 days post treatment follow-up period, and he/she considers there is a reasonable possibility that the event is causally related to the study treatment, the investigator should notify AstraZeneca, Patient Safety by reporting the SAE via both the eCRF in Medidata Rave and paper SAE report to AstraZeneca DES.

At any time after a patient has completed the study, if an investigator learns of any SAE including sudden death of unknown cause, and there is a reasonable possibility that the event is causally related to the investigational product, this should be notified to AstraZeneca, Patient Safety. Otherwise, after study treatment completion (i.e. after any scheduled post treatment follow-up period has ended) there is no obligation to actively report information on new AEs or SAEs occurring in study patients. This includes new AEs/SAEs in patients still being followed up for survival but who have completed the post treatment follow up period (30 days).

Any case of MDS/AML or new primary malignancy occurring at any time from signature of informed consent for the entire participation of the patient in the study including the follow-up period should be reported as an SAE. Any MDS/AML, new primary malignancies or pneumonitis occurring after the 30 day follow up period should be reported to AstraZeneca Patient Safety regardless of causality, investigator's assessment or knowledge of treatment arm. Non-melanoma skin cancers need to be reported as a non-serious AE unless at least one of the seriousness criteria is met and then it must be reported as an SAE, see Section 6.4.2 of the CSP. Any of these type of serious or non-serious events need to be reported to AstraZeneca Patient Safety according to SAE reporting procedures for this study, regardless of investigator's assessment of causality or knowledge of the treatment arm. If a patient develops MDS/AML full diagnostic details and classification should be provided e.g. bone marrow and cytogenetic analysis reports, see Sections 5.5.6.3 and 6.4.5.5 of the CSP. A questionnaire will be sent to any investigator reporting MDS/AML or new primary malignancy so that relevant details can be reported.

\*In Screening PART 1 of the study only SAEs related to study mandated procedures (i.e. blood draw) will be collected. In Screening PART 2 all SAEs will be collected.

#### 3.3.1.1 Olaparib adverse events of special interest (AESI)

Adverse events of special interest (AESI) are events of scientific and medical interest specific to the further understanding of olaparib's safety profile and require close monitoring and rapid communication by the investigators to AstraZeneca. Adverse events of special interest for olaparib are MDS/AML, new primary malignancy (other than MDS/AML) and pneumonitis. The search strategy to identify AESIs as provided by AstraZeneca Patient Safety is shown in Table 6.

Table 6 Search strategy to identify AESI

| MDS/AML | Myelodysplastic syndrome (SMQ-Narrow) +AML PTs: Acute biphenotypic leukaemia, acute leukaemia, acute megakaryocytic leukaemia, acute monocytic leukaemia, acute myeloid leukaemia, acute myeloid leukaemia recurrent, acute myelomonocytic leukaemia, acute promyelocytic leukaemia, acute undifferentiated leukaemia, blast cell crisis, blast crisis in myelogenous leukaemia, chloroma, eosinophilic leukaemia, erythroleukaemia, leukaemia basophilic, leukaemia granulocytic, leukaemia monocytic, myeloid leukaemia, |
|---|---|
| | transformation to acute myeloid leukaemia |
| Other NPMs | Malignant or unspecified tumours (SMQ) |
| Pneumonitis | Interstitial Lung Disease (SMQ-Narrow) |

Note: this search strategy could be updated at any point up to database lock.

#### 3.3.2 Treatment exposure

Exposure will be defined as follows:

#### Total (or intended) exposure of olaparib/placebo

• Total (or intended) exposure (days) = last dose date - first dose date + 1

Last dose date is defined as earliest of:

- Last dose date at discontinuation
- Last dose date at treatment completion
- Last dose date at Data cut off (DCO)

#### Actual exposure of olaparib/placebo

• Actual exposure (days) = Total exposure – Total duration of dose interruptions, where Total exposure will be calculated as above.
### Number of days on 300 mg olaparib/placebo bd.

• Number of days on 300 mg olaparib/placebo bd. = actual exposure for the dose assigned.

# **Cumulative exposure**

Cumulative exposure over time is categorized by duration of total intended exposure in months of cumulative exposure;>0 months,  $\geq$  1 month,  $\geq$  2 months,  $\geq$  3 months,  $\geq$  4 months,  $\geq$  5 months,  $\geq$  6 months,  $\geq$  7 months,  $\geq$  8 months,  $\geq$  9 months,  $\geq$  10 months,  $\geq$  11 months, 12 months. Subjects are counted under each category providing their total intended exposure is up to and including that duration.

# Exposure by dose

The following summaries are produced for exposure by dose;

- Range of any dose for any subject = minimum dose for any subject (mg/day) -maximum dose for any subject (mg/day)
- Mean dose (mg/day) = mean (any dose (mg/day) for any subject)
- Range of mean doses = minimum (mean dose (mg/day) per subject) maximum (mean dose (mg/day) per subject)
- Mean total cumulative dose (mg) = mean (cumulative dose (mg) per subject)
- Range of total cumulative doses (mg) = minimum (cumulative dose (mg) per subject) maximum (cumulative dose (mg) per subject)
- Range of maximum doses = minimum (maximum dose (mg/day) per subject) maximum (maximum dose (mg/day) per subject)

# Olaparib total daily dose

The total daily dose is defined as the mean total daily dose for each subject in each 3 month period.

- $>500 \text{ to } \le 600$
- >400 to <500
- <400

Over three monthly periods

- Up to 3 months
- >3 to  $\leq$ =6 months
- >6 to <=9 months
- >9 to <=12 months

In each time period the total daily dose for each patient is as shown in the categories above, the number and % of patients with total daily dose as categorised will be presented, the denominator is the number of patients receiving Olaparib in that time period.

Appendix C gives an example of how to consider patients who permanently discontinued treatment during a dose interruption.

# 3.3.3 Dose intensity

Relative dose intensity (RDI) is the percentage of the actual total dose delivered relative to the intended total dose through to treatment discontinuation. Percentage intended dose (PID) is the percentage of the actual total dose delivered relative to the intended total dose through to invasive disease recurrence. Both will be derived using study treatment data up to one year or until the date of invasive disease (whichever is earliest).

Relative dose intensity (RDI) and percent intended dose (PID) will be defined as follows:

• RDI = 100% \* d/D, where d is the total actual dose delivered up to the earlier of a censoring event or the actual last day of dosing and D is the total intended dose up to a censoring event or the actual last day of dosing. The censoring events are Trinvasive disease, withdrawal from study and DCO.

For example: For a patient with a date of invasive disease before the date of last study treatment, the date of invasive disease is treated as a censoring event, i.e. the total intended dose (D) is calculated until the date of recurrence.

• PID = 100% \* d/D, where d is the total actual dose delivered up to invasive disease or a censoring event or the actual last day of dosing and D is the total intended dose up to invasive disease or a censoring event. The censoring events are withdrawal from study and DCO. D is the total dose that would be delivered, if there were no modification to dose or schedule.

Due to the eCRF design, the actual cumulative dose does not capture all missed or forgotten doses within an individual day. This will be recorded as if the patient took a full daily dose, which could lead to an overestimation of RDI and PID.

Examples of calculating RDI and PID are given in Appendix C.

### 3.3.4 Laboratory data

Laboratory data will be collected throughout the study, from screening to follow-up visit as described in Table 1 and Table 2 of the CSP. Blood and urine samples for determination of haematology, clinical chemistry, and urinalysis will be collected as described in Section 6.4.5 of the CSP.

### 3.3.5 ECGs

ECGs are required during screening within 28 days prior to randomisation and when clinically indicated afterwards. All ECGs should be assessed by the investigator as to whether they are clinically significantly abnormal / not clinically significantly abnormal.

# 3.3.6 Vital signs

Vital signs data obtained up until the 30 days from date of last dose of olaparib/placebo treatment will be used for reporting. For derivation of post baseline visit values considering visit window and to handle multiple records, derivation rules as described in Section 3.3.7 below will be used.

# 3.3.7 General consideration for safety assessments

Time windows will be defined for any presentations that summarise values by visit (see below). The following conventions should also apply:

- The time windows should be exhaustive so that data recorded at any time point has the potential to be summarised. Inclusion within the time window should be based on the actual date and not the intended date of the visit.
- All unscheduled visit data should have the potential to be included in the summaries.
- The window for the visits following baseline will be constructed in a way that the upper limit of the interval falls half way between the two visits (the lower limit of the first post-baseline visit will be Day 2). If an even number of days exists between two consecutive visits then the upper limit will be taken as the midpoint value minus 1 day.

For example, the visit windows for laboratory data are:

- Week 2, Day 15, visit window 2 21
- Week 4, Day 29, visit window 22 42
- Week 8, Day 57, visit window 43 70
- − Week 12, Day 85, visit window 71 98
- Week 16, Day 113, visit window 99 126
- Week 20, Day 141, visit window 127 154
- Week 24, Day 169, visit window 155 217
- Week 38, Day 267, visit window 218 315
- Week 52, Day 365, visit window 316 379

- For summaries showing the maximum or minimum values, the maximum/minimum value recorded on treatment will be used (regardless of where it falls in an interval).
- Listings should display all values contributing to a time point for a patient.
- For visit based summaries:
  - If there is more than one value per patient within a time window, then the
    closest value should be summarised, or the earlier in the event the values
    are equidistant from the nominal visit date. The listings should highlight
    the value for that patient that went into the summary table, wherever
    feasible.
  - To prevent the creation of very large tables or plots that contain many cells with meaningless data, the visit data for each treatment group should only be summarised if the number of observations is greater than the minimum of 20 and > 1/3 of patients dosed.
- For summaries at a patient level, all values should be included, regardless of whether they appear in a corresponding visit based summary, when deriving a patient level statistic e.g. a maximum.
- Baseline will be defined as the last non-missing measurement prior to dosing with study treatment (olaparib or placebo). For laboratory data and vital signs data, any assessments made on day 1 will be considered pre-dose. Where safety data are summarised over time, study day will be calculated in relation to date of first treatment (olaparib or placebo).

Missing safety data will generally not be imputed, although partial/missing start and end dates for adverse events and concomitant medications will be imputed (see Section 4.2.15). However, safety assessment values of the form of "< x" (i.e., below the lower limit of quantification) or > x (i.e., above the upper limit of quantification) will be imputed as "x" in the calculation of summary statistics but displayed as "< x" or "> x" in the listings.

# 3.3.8 PK variables

The PK and PKPD analysis will be described in detail in a separate modelling analysis plan.

Pharmacokinetic (PK) sampling will be performed in a subset of patients. Each patient will be asked to contribute 5 blood samples, one from each of the predefined time windows below preferably on visit 4, day 29. Nevertheless, the samples can also be taken at a later treatment visit, provided that PK consent was obtained beforehand.

- Pre-dose (before morning dose)
- Between 0 and 0.5 hour post-dose
- Between >0.5 and 1.5 hour post-dose
- Between 3 and 6 hours post-dose
- Between >6 and 12 hours post-dose (before evening dose).

The PK analysis of the plasma concentration data for olaparib will be performed by Covance on behalf of Clinical Bioanalysis Alliance, AstraZeneca R&D, using an appropriate bioanalytical method. The actual sampling times will be used in the PK calculations. For each patient providing a complete set of PK samples, non-linear mixed effects modelling (NONMEM) will be used to estimate steady state  $C_{max}$ , AUC and  $C_{min}$ .

# 3.4 Resource use

Resource use for serious adverse events (including hospitalisations) will be captured through the serious adverse events reporting procedures.

Resource use outcome variables include the following:

- Length of hospital stay
- Number of hospital admissions

The length of hospital stay will be calculated as the difference between the date of hospital discharge (or death date) and the start date of hospitalisation or start of study drug if the start of study drug is after start date of hospitalisation (length of hospital stay = end date of hospitalisation – start date of hospitalisation + 1). Patients with missing discharge dates will be calculated as the difference between the last day with available data and the start date of hospitalisation.

Sum of total duration of hospital stay will be considered for analysis if patient was admitted to hospital more than one time during study period.

### 4. ANALYSIS METHODS

The primary analysis of IDFS will occur when 330 IDFS events have occurred (have been counted in the clinical database).

An initial analysis of OS and DDFS will be performed at the same time as the primary analysis of IDFS and will use the same methodology and model.

The final OS analysis will be conducted once the trial follow up is complete (i.e. 10 years from when the last patient is randomised, estimated 15 years from first patient randomised assuming recruitment of 5 years).

In addition, an analysis will be performed half way between the primary IDFS analysis and the final overall survival analysis (estimated around 10 years from first patient randomised but timings will be driven by the primary IDFS analysis once known). At this time point both DDFS and OS will be analysed and some alpha (see Section 5 for full details) will be reserved for formal hypothesis testing. IDFS may also be updated if more information is available but this would be considered a supportive update of the primary analysis and no alpha will be reserved for IDFS.

For details on alpha spend and how this will be allocated across the planned analyses, see Section 5

Supportive analyses of contralateral invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer will be provided at the interim and at the primary analysis of IDFS, however no multiple adjustment will be applied as these are viewed as supportive endpoints.

# 4.1 General principles

The primary statistical analysis of the efficacy of olaparib will include all randomised patients and will compare the treatment groups on the basis of randomised treatment, regardless of the treatment actually received. Patients who were randomised but did not subsequently go on to receive study treatment are included in the Full Analysis Set. Therefore, all efficacy will be summarised and analysed in the FAS on an intention-to-treat basis. All patient reported outcome data will be summarised and analysed in a subset of the FAS, the PRO analysis set.

When assessing safety and tolerability, summaries will be produced based on the Safety Analysis Set. This will include all patients who receive at least one dose of randomised treatment (olaparib or placebo). Patients in the Safety Analysis Set will be analysed by whether or not the patient received at least one dose of olaparib. The safety data will be summarised descriptively and will not be formally analysed.

If there are any randomised patients not confirmed to have a *gBRCA* mutation by the central test, a subset of confirmed gBRCAm patients will be defined for sensitivity analyses. In this case, key efficacy, demographic, patient characteristics and safety outputs will be repeated in this subset.

Summary statistics for continuous variables will include the number of subjects, mean, standard deviation, median, minimum, and maximum values. Continuous variables will generally be presented with the mean and median to 1 decimal more than the individual data, and the standard deviation to 2 decimals more than the individual data. Summary statistics for categorical variables will include frequencies and percentages. Percentages will be presented to one decimal place.

The SAS programming language will be used to produce all outputs except for the test of non-proportional hazards by Grambsch-Therneau methods. This analysis will use the R package survival (Therneau and Grambsch 2000; Therneau 2015), specifically the coxph (Therneau and Grambsch 2000) and cox.zph (Grambsch and Therneau 1994) functions.

A SAS macro for the GailSimon method will be used (see appendix D).

# 4.2 Analysis methods

The treatment comparison is olaparib 300 mg bd. versus placebo.

If the significance level has been adjusted for an analysis (e.g. interim analysis of IDFS) then results will be presented using a confidence interval corresponding to the significance level applied and a 95% CI will also be presented for descriptive purposes. Otherwise, results of all statistical analysis will be presented using a 95% CI. All p-values presented will be 2-sided.

# 4.2.1 Confidence intervals at the interim analysis

In the event of stopping for efficacy at the interim analysis the secondary endpoints will be analysed according to the rules in Section 5 Interim Analyses: 4% on DDFS and 1% on OS, inferential and exploratory CIs will be reported for DDFS and OS.

Inferential confidence intervals will be presented for IDFS, and, if the null is rejected for IDFS, they will also be presented for OS and DDFS.

Under the scenario of no alpha recycling (i.e. both OS and DDFS rejected or accepted) the following intervals will be presented;

IDFS: 99.5%DDFS: 99.5%OS: 99.8%

If the null is rejected for OS and not for DDFS then alpha will be recycled to DDFS from OS. In this scenario the following intervals will be presented;

IDFS: 99.5%DDFS: 99.375%OS: 99.8%

If the null is rejected for DDFS and not for OS then alpha will be recycled to OS from DDFS. In this scenario the following intervals will be presented;

IDFS: 99.5%DDFS: 99.5%OS: 99%

# 4.2.2 Median clinical follow-up

Median clinical follow-up will be calculated using the reverse censoring method (Schuster, 1991; Schemper, 1996)

# 4.2.3 Kaplan-Meier estimates of IDFS

IDFS times will be summarized using Kaplan-Meier survival curves (Kaplan & Meier, 1958).

### 4.2.4 Percentages of invasive disease free subjects at yearly intervals

The percentages of surviving subjects who are invasive disease free at yearly intervals from the time of randomisation will be estimated from the Kaplan-Meier curves (Kaplan & Meier,

1958). This will include at a minimum the following time points as the data become available during the trial: 1 year, 2 years, and 3 years. Approximate 95% confidence limits will be calculated, based on Greenwood's formula (Collett 2003) for the standard error of the Kaplan-Meier estimate

The following table details which endpoints are to be subject to formal statistical analysis.

Table 7 Formal Statistical Analyses to be Conducted

| Endpoints Analysed | Notes |
|---|---|
| IDFS (Time from randomisation to invasive disease recurrence or death due to any cause) | Primary analysis stratified log-rank test and Cox regression |
| | Key sensitivity analysis: Stratified Cox regression in randomised patients confirmed as gBRCA mutation positive by central test (if different from FAS(ITT)) |
| Overall Survival (Time from randomisation to death due to any cause) | Stratified log-rank test and Cox regression |
| | Key sensitivity analysis: Stratified Cox regression in randomised patients confirmed as gBRCA mutation positive by central test (if different from FAS(ITT)) |
| DDFS (Time from randomisation to distant recurrence or death due to any cause) | Stratified log-rank test and Cox regression |
| | Key sensitivity analysis: Stratified Cox regression in randomised patients confirmed as gBRCA mutation positive by central test (if different from FAS(ITT)) |
| Incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, primary fallopian tube cancer and new primary peritoneal cancer | Fine and Gray models |
| FACIT-Fatigue | Primary analysis MMRM at 6 and 12 months |
| | Sensitivity analysis MMRM |
| EORTC QLQ-C30 GI symptoms | MMRM |
| EORTC QLQ-C30 HRQoL | MMRM |

### 4.2.5 Demographic and baseline characteristics data

The following will be summarised by randomised treatment group:

- Patient disposition
- Important deviations
- Inclusion in analysis populations
- Demographics (age, age group, sex, race and ethnicity)
- Patient characteristics at baseline (height, weight, weight group, body mass index (BMI) and BMI group)
- Stratification factors recorded on the eCRF
- Stratification factors according to the randomisation system.
- Local and central BRCA mutation type (using the central PMG)
- Breast cancer surgical history (breast conservation; sentinel nodal status; axillary nodal status)

The following will be summarised by randomised treatment group:

- Patient recruitment by country and centre
- Receptor status (HER2 status, ER status, PgR status) from local and central
- Prior chemotherapy for primary breast cancer and for primary malignancies (including anthracycline, taxane, and anthracycline plus taxane)
- Prior hormone therapy for primary breast cancer and for primary malignancies
- Prior platinum therapy for primary breast cancer and for primary malignancies
- Pathological characteristics of primary breast cancer at baseline (bilateral, histological grade, clinical stage and pathological stage, CPS+EG score)
- ECOG performance status at baseline
- Ovarian surgical history (both ovaries removed: Yes; No) Note: oophorectomy is collected on the Procedures eCRF page
- Fallopian tube surgical history (Note: salpingectomy is collected on the Procedures eCRF page
- Time from last treatment (surgery, chemotherapy or radiotherapy) to randomisation
- Time from diagnosis to randomisation
- Medical History
- Disallowed concomitant medications
- Allowed concomitant medications
- Post-discontinuation disease-related cancer therapy
- Post-event treatments/radiotherapy/surgery
- Family history of cancer

For concomitant medication coding the WHO Drug Dictionary Enhanced with Herbal Dictionary (release date 1st March 2016)

Prior chemotherapy, platinum therapy, primary breast cancer surgery and ovarian surgery will also be summarised separately for patients who received neo-adjuvant or adjuvant chemotherapy, and pathological characteristics will be summarised according to hormone receptor status and neo-adjuvant or adjuvant chemotherapy. In addition, prior and/or concurrent hormone therapy will be summarised separately for ER and/or PgR positive /HER2 negative patients.

The total number of patients unblinded and patients who were unblinded (a) prior to invasive disease recurrence and (b) prior to or on the day of treatment discontinuation will be summarised by treatment group.

Patient disposition, demographic and patient characteristics, and pathological characteristics will also be presented in the confirmed gBRCAm patients if appropriate.

# 4.2.6 Multiplicity

The primary endpoint of the study is IDFS. However, key secondary endpoints will be OS and DDFS.

In order to describe the nature of the effects of olaparib treatment IDFS, DDFS and OS will be tested at a 2-sided significance level of 5%. However, in addition, in order to strongly control the overall type I error at 2.5% 1-sided (5% 2 sided), a multiple testing procedure (MTP) will be employed across the primary endpoint and all key secondary endpoints intended for label claims (DDFS and OS). The MTP will account for any interim analyses on IDFS, DDFS and OS and also planned further analyses post the primary 330 IDFS event data cut off.

A hierarchical testing strategy will be employed where IDFS is tested first using the full test mass (i.e. full 2.5%, 1-sided alpha), then DDFS and OS will be tested if IDFS is significant based on a weighted proportion of the test mass (2% for DDFS and 0.5% for OS, 1-sided) which can be recycled to secondary endpoints not yet rejected. Testing stops when the entire test mass is allocated to non-rejected endpoints.

Figure 3 Multiple Testing Procedure



IDFS is planned to be analysed at the interim and the final analysis (see Section 5 for further details). If IDFS is significant at the interim based on the ITT population then secondary endpoints will be formally tested at the interim based on the MTP outlined above. To account for multiple analyses on each endpoint a separate alpha spending function will be applied to each endpoint (Glimm et al 2009). Further analyses of DDFS and OS with more mature follow-up may be required for which some alpha will be reserved for significance testing.

All planned analyses will be performed, regardless of the outcome of the MTP. If the full test mass has been used on an earlier test in the MTP, no claims regarding the statistical significance of a subsequent analysis in the MTP will be made.

# 4.2.7 Primary endpoint - Invasive Disease-Free Survival (IDFS)

# 4.2.7.1 Primary Analysis

As described in Section 3.1.1, patients who have not had a recorded IDFS event at the time of the analysis will be censored at the date of last contact if lost to follow-up or withdrawn from study or their last disease evaluation if follow-up is ongoing.

Patients will be censored at 0.5 days after randomisation under the following 3 circumstances:

- Patients who have had an event prior to randomisation.
- Patients who were identified as inadvertent randomisations (i.e. patient was randomised and the site later realised that they should not have been randomised, they have had no follow-up nor did they receive treatment).
- Patients who have withdrawn consent, received no treatment, and will not be providing any follow-up data.

These randomised patients will be counted in the Full Analysis Set, however they will be treated as being censored for the IDFS event just after randomisation. Censoring these patients at day 0.5 will not affect the log-rank test, however, they will be counted in the total number at risk and in the Kaplan-Meier (KM) plot. The reason for censoring at day 0.5 is to avoid ties with other patients censored on day 1.

IDFS will be analysed using a log-rank test stratified by the stratification factors (using the information entered into the randomisation system) and the corresponding p-value will be reported as the primary analysis result.

In addition, IDFS will be analysed using a stratified Cox proportional hazard model incorporating the Efron approach for handling ties. As with the IDFS analysis, the stratification factor categories used in the Cox model will be those identified for each patient at the time of randomisation. The point estimate of the treatment effect, i.e., the hazard ratio of IDFS (olaparib vs. placebo) will be obtained by maximizing the Cox partial likelihood function, which is the product of the partial likelihood of each stratum. The 95% confidence interval will be estimated using the profile likelihood approach. Should the conclusion from the log-rank test not agree with the score test from the Cox proportional hazards model, the log-rank test will dominate.

A KM plot of IDFS, with tick marks to identify censored observations, will be presented by treatment group. Summaries of the number and percentage of patients experiencing an IDFS event, and the site of first event (see Section 3.1.1 for the hierarchy) will be provided for each treatment group.

The estimated 3 year IDFS will be summarised (using estimates from the KM curve) and presented by treatment group.

The primary stratified log-rank test of IDFS will be based on the stratification factors determined from the following pooling strategy.

In the event that there are fewer than 5 IDFS events per treatment arm within any individual stratum (initially starting with 16 strata; 16=2x2x2x2 including treatment group), one stratification factor will be removed at a time until there are at least 5 IDFS events within each individual stratum in the following order:

- 1 Prior platinum use for breast cancer (yes/no)
- 2 Prior chemotherapy (neo-adjuvant vs. adjuvant)
- 3 Hormone receptor status (ER and/or PgR positive/HER2 negative vs. TNBC)

The additional Cox analysis will be based on the same stratification factors. An unadjusted analysis will also be done as a sensitivity analysis and compared with the primary results.

### 4.2.7.2 Sensitivity Analyses for IDFS

The following sensitivity analyses will be done to compare against the primary IDFS analysis result. For each of the analyses specified the HR and CI from the Cox model will be reported alongside. The stratification factors for the sensitivity analyses will be the same as for the main analysis with the exception of the unadjusted analysis, mis-stratification in the randomisation system and the central pathology review, stratification factors for these are detailed below.

# If applicable, an analysis will be performed for IDFS using the same model as described above but based on all randomised patients confirmed to have *gBRCA* mutations by the central test. This analysis is only required if the analysis population differs from the primary ITT population (i.e. only required if any of the randomised patients are not confirmed to have *gBRCA* mutations by the central test).

# Mis-stratification in the randomisation system

Any patients mis-stratified in the randomisation system (i.e. incorrect details are entered at the time of randomisation) will be included in the primary analysis as stratified. Cross-tabulations of stratification factors from the randomisation system and the correct baseline data from the eCRF will be considered. If >5% of randomised patients are incorrectly stratified (i.e. randomisation system data does not match baseline data) then a sensitivity analysis will be performed for IDFS using the same model as described above but using the eCRF information.

Stratification factors and therefore the stratification errors will be based on the pooling strategy identified for the main IDFS analysis. For example, if only HR status is a stratification factor following the pooling for the main IDFS analysis then only the stratification errors between HR status on the randomisation system and on the eCRF will be taken into account when calculating the % of stratification errors. Under this scenario, if the sensitivity analysis was triggered then it would only include HR status from the eCRF as a stratification factor in the fitted Cox model.

### Central pathology review

If the results of ER and PgR status from the local and central labs differ in >5% of randomised patients, then a sensitivity analysis will be performed for IDFS using the same model as described above, but using the central lab result to determine the HR status stratification factor and compared with the primary analysis result.

Note: central HR status results not available for China.

### **Important PDs**

A 'deviation bias' sensitivity analysis may be performed excluding patients with IPD's that may affect the efficacy of the trial therapy. Further details are given in Section 2.2.

### Unadjusted analysis

An unadjusted (unstratified Cox model) analysis will be performed as a sensitivity analysis and compared with the primary results.

### **Assumption of proportional hazards**

The assumption of proportional hazards underlying the log-rank test and the Cox model used for the primary analysis will be assessed. Proportionality will be assessed using two approaches, firstly by inspecting plots of complementary log-log (time) versus log (time) and secondly by formally testing using the Grambsch–Therneau test (G-T) based on scaled Schoenfeld residuals from a Cox model including treatment group as a factor. If the G-T test is significant (p<0.05), and proportionality is rejected, Restricted Mean Survival Time (RMST) methods will be used to estimate and test the treatment difference while allowing for non-proportional hazards. RMST will be based on the Pseudo-observations method (Anderson et al 2004) with covariates included in the model using Generalised estimating equations (GEE) with robust standard errors.

The cut-off time (t\*) for RMST will be the minimum of the largest observed event time over the two treatment groups. Note: in the presence of non-proportionality, the HR point estimate of the treatment difference obtained from the main analysis of the IDFS primary end-point (in Section 4.2.3.1) will be interpreted as an average HR over the observed extent of follow-up. Note: in the presence of non-proportionality, the HR will be interpreted as an average HR over the observed extent of follow-up.

As described in Section 3.3.1, patients with events prior to randomisation will be censored at 0.5 days after randomisation. In addition, the IDFS analysis will be run excluding these patients from the Full Analysis Set.

# **Interval censored Cox regression**

A sensitivity analysis will be performed where patients whose visit schedule has not been according to the protocol are fitted in the Cox model using interval censoring.

### Specifically;

- For patients experiencing an event, and without follow-up according to the protocol (defined as over 18 months between the event and the last visit), the interval from the last date at which the subject was known to be IDFS free to the date of recurrence or death, will be used.
- For patients that were previously censored, or had an event and were seen according to the protocol defined visit schedule, the lower limit of the interval will be set to the censoring/event date, while the upper limit will be set to missing.

Note: Missed visit will be defined according to the year of study that a patient is in, and incorporate the allowed windows.

This analysis will be performed using SAS function PROC ICLIFETEST. The ICLIFETEST procedure performs nonparametric survival analysis for interval-censored data. Default weight function will be used, this is the generalised log-rank test with constant weights over time.

# 4.2.7.3 Subgroup analyses

Subgroup analyses will be conducted to assess consistency of treatment effect across potential or expected prognostic factors, including the baseline stratification factors determined from the eCRF data

The interaction between treatment and subgroup will be assessed by fitting an unstratified Cox model with the two main effects; treatment and subgroup, with the interaction term for treatment by subgroup.

Patients with missing data for subgroups will not be included in the subgroup analysis.

Hazard ratios will not be presented for any subgroup levels with less than 5 events in either treatment arm. The HAZARDRATIO statement in the PHREG procedure in SAS will only include levels with at least 5 events in both treatment arms.

For example: subgroup analysis for BRCA gene name has 3 levels

- BRCA1
- BRCA2
- BRCA1/2

If subgroup levels for BRCA1 and BRCA2 have at least 5 events in both treatment arms, and there are less than 5 events in either one of the BRCA1/2 treatment arms then the patients associated with subgroup BRCA1/2 will still be included in the analysis as the level provides valuable information, however the hazard ratio will not be generated.

The following subgroups are of primary interest:

• Neoadjuvant chemotherapy; adjuvant chemotherapy

This will be determined from the response to the variable "Intent" (prior neo-/adjuvant chemotherapy for primary breast cancer page) on the eCRF at randomisation.

Note: a patient should only have either prior adjuvant chemotherapy or prior neoadjuvant chemotherapy and no patient should have received both. Patients for whom it is not possible to determine their chemotherapy "intent" from the CRF, will be categorised according to how they were randomised.

Prior chemotherapy will be coded for the analysis as follows

- 0= Prior neoadjuvant chemotherapy
- 1= Prior adjuvant chemotherapy
- Prior platinum therapy for current breast cancer (Yes; No)

This will be determined from the WHODrug coded term associated with response to the variable "Treatment name" (prior neo-/adjuvant chemotherapy for primary breast cancer page) on the eCRF at randomisation. If the coded term is 'Platinum compound, the patients will be considered a "Yes". Otherwise, they will be considered a "No".

Prior platinum therapy will be coded for the analysis as follows

- 0= No
- 1= Yes
- Hormone receptor status (ER and/or PgR positive /HER2 negative; TNBC)

ER status will be determined from the response to "ER status" and PgR status will be determined from the response to "PgR status" (local laboratory page; hormone receptor status section) on the eCRF at randomisation.

- 0= ER and/or PgR positive/HER2 negative
- 1= TNBC
- BRCA mutation type (BRCA1, BRCA2 or BRCA1/2 both)

This will be determined from the BRCA mutation type based on central data.

- 0=BRCA1
- 1=BRCA2
- 2=BRCA1/2 both
- Hormone receptor status by prior chemotherapy setting
  - 0= ER and/or PgR positive with neoadjuvant chemotherapy
  - 1= ER and/or PgR positive with adjuvant chemotherapy
  - 2= ER and PgR negative with neoadjuvant chemotherapy

- 3= ER and PgR negative with adjuvant chemotherapy
- BRCA status by prior platinum therapy setting
  - 0=BRCA1 with prior platinum therapy for current breast cancer
  - 1=BRCA1 with no prior platinum therapy for current breast cancer
  - 2=BRCA2 with prior platinum therapy for current breast cancer
  - 3=BRCA2 with no prior platinum therapy for current breast cancer
  - 4=BRCA1/2 both with prior platinum therapy for current breast cancer
  - 5=BRCA1/2 both with no prior platinum therapy for current breast cancer

The following additional subgroups will also be analysed to assess consistency in treatment effect across a broader set of baseline characteristics known before start of study medication:

• Type of prior Neoadjuvant/Adjuvant chemotherapy (anthracycline; taxane; anthracycline plus taxane)

This will be determined from the WHODrug coded term associated with response to "Treatment name" from the prior neo-/adjuvant chemotherapy for primary breast cancer page on the eCRF at randomisation. The following therapies will be considered to each category

- 0= Prior anthracycline alone
- 1=Prior taxane alone
- 2= Prior anthracycline and taxane
- Type of breast surgery prior to randomisation (breast conservation; unilateral mastectomy)

This will be determined from the response to "Type of surgery" (Breast cancer surgery page; primary breast cancer surgery section) on the eCRF at randomisation.

- 0= Breast conservation defined as Partial mastectomy / Breast Quadrantectomy
   / Breast Segmentectomy / Breast Lumpectomy and Breast re-excision of margins
- 1= unilateral mastectomy defined as Modified radical mastectomy, Radical mastectomy (Halsted) or Simple mastectomy
- 2= bilateral mastectomy defined as Bilateral Mastectomy

• Have both ovaries been removed? (Yes; No)

This will be determined from the Procedures page on the eCRF and will only include ovarian surgeries prior to the first dose of study medication. Note: if the number of patients with local mastectomy/ oophorectomy or bilateral mastectomy/ oophorectomy is low then local and bilateral may be combined into one category.

- 0= not bilateral oophorectomy
- 1= bilateral oophorectomy
- Axillary nodal status at surgery prior to randomisation: (Positive or negative for the TNBC, adjuvant patients only)

This will be determined from the response to "Axillary sentinel node biopsy" (breast cancer surgery page; sentinel node sampling section) on the eCRF at randomisation.

- 0= node negative
- 1= node positive
- CPS+EG score at baseline (2, 3 or 4; 5 or 6 for the post neoadjuvant group only)

This will be derived from the responses to "CPS &EG Score" on the Breast Cancer History Form. These scores are checked by data management.

- 0= CPS+EG score of 2, 3 or 4
- 1= CPS+EG score of 5 or 6
- Age at randomisation (<50; 50-64;  $\ge 65$ )

This will be determined from "AGE at randomisation" which is derived in the database using the patient's date of birth (informed consent and demography page). The following categories may be revised after consideration of the distribution of ages when recruitment has been completed.

- 0= Age < 50 years
- 1= Age 50 64 years
- 2= Age ≥65 years
- Race (White, Black/African-American, Asian and Other [Native Hawaiian/Pacific Islander or American Indian/Alaska Native or Others])

This will be determined from the response to "Race" (informed consent and demography page) on the eCRF at Randomisation. Note: from the study schedule (Table 2) that Race data will be collected unless not allowed by local regulations.

- 0= White
- 1= Black/African-American
- 3=Asian
- 4=Other
- Ethnicity (Hispanic or Latino; Not Hispanic or Latino; Not known, not recorded or refused)

This will be determined from the response to "Ethnicity" (informed consent and demography page) on the eCRF at Randomisation. Note: from the study schedule (Table 2) that Ethnicity data will be collected unless not allowed by local regulations.

- 0= Hispanic or Latino
- 1= Not Hispanic or Latino
- 2=Not known, not recorded or refused
- Jewish descent (Ashkenazi Jewish descent or not of Ashkenazi Jewish descent)

This will be determined from the response to question on Jewish descent (informed consent and demography page) on the eCRF at Randomisation.

- 0= Not of Ashkenazi Jewish descent
- 1= Yes, of Ashkenazi Jewish descent
- Sponsor (AZ; NRG)

This will be determined from the centre number.

- 0 = AstraZeneca (AZ)
- 1 = NRG
- Geographic region
  - 0= North America (Canada, United States of America)

- 1= South America (Argentina, Brazil, Chile, Colombia, Costa Rica, Guatemala, Mexico, Panama, Peru, Philippines, Puerto Rico, Uruguay, Venezuela)
- 2= Europe (Austria, Belgium, Bulgaria, Croatia, Czech Republic, Denmark, Estonia, Finland, France, Georgia, Germany, Great Britain, Greece, Hungary, Iceland, Ireland, Italy, Latvia, Lithuania, Luxembourg, Netherlands, Norway, Poland, Portugal, Romania, Russian Federation, Serbia and Montenegro, Slovakia, Slovenia, Spain, Sweden, Switzerland, Turkey, Ukraine)
- 3= Asia Pacific and South Africa (Afghanistan, Australia, China, Hong Kong, India, Indonesia, Israel, Japan, Malaysia, New Zealand, South Korea, Singapore, South Africa, Taiwan, Thailand, Vietnam)

Other baseline variables may also be assessed if there is clinical justification.

To avoid potential problems with non-proportionality in the covariates, the HRs (olaparib: placebo) and profile likelihood CIs for the treatment effect will be calculated from a Cox proportional hazards model (using the Efron approach for handling ties) for each level of the subgroup. The model will include factors for treatment group and subgroup and the treatment-by-subgroup interaction. All patients with non-missing subgroup data will be included in the model. However, HR/CI estimates from the model will only be displayed in categories with sufficient number of events available (at least 5 events in both treatment groups). For subgroups with too few events we will only display the number of patients and number (%) of events.

For subgroups with sufficient number of events, we will display all stats including the HR/CI estimates from the model in a table. In addition, the HRs and 95% CIs will be presented on a forest plot including the HR and 95% CI from the overall population (using the primary analysis). The p-value for interaction TRT\*SUBG will also be presented, to be assessed at a 10% level for the purpose of hypothesis generation.

No adjustment to the significance level for testing subgroups will be made since all these subgroup analyses will be considered exploratory. The results would be used as supportive data for the primary analysis of IDFS based on all randomised patients.

For each subgroup, a Kaplan-Meier plot of IDFS, with tick marks to identify censored observations, will be presented by treatment group and summaries of the IDFS survival probabilities for each treatment will also be produced.

### 4.2.7.4 Analysis of interactions

The presence of quantitative interactions will be assessed by means of an overall global interaction test. This will be performed in the overall population by comparing the fit of a Cox proportional hazards model including treatment, all covariates (including stratification factors as derived from the eCRF data), and all covariate-by-treatment interaction terms, with one that excludes the interaction terms and will be assessed at the 2-sided 10% significance level.

Plausible covariates include only the stratification factors, therefore the full model fitted will include the 3 stratification factors and treatment as main effects, and the two way interactions between each stratification factor and treatment.

If a covariate does not have at least 20 events per level (of the covariate) it will be included as a covariate in the model, but the covariate-by-treatment interaction term will be omitted. If the fit of the model is not significantly improved then it will be concluded that overall the treatment effect is consistent across the subgroups.

If the global interaction test is found to be statistically significant, an attempt to determine the cause and type of interaction will be made. Stepwise backwards selection will be performed on the full model, whereby (using a 10% level throughout) the least significant interaction terms are removed one-by-one and any newly significant interactions re-included until a final model is reached where all included interactions are significant and all excluded interactions are non-significant. Throughout this process all main effects will be included in the model regardless of whether the corresponding interaction term is still present. This approach will identify the factors that independently alter the treatment effect and prevent identification of multiple correlated interactions.

Any quantitative interactions identified using this procedure will then be tested to rule out any qualitative interaction using the approach of Gail and Simon 1985. This will be done using SAS macro %GailSimon (Appendix D).

# 4.2.8 Overall survival (OS) and Distant disease free survival (DDFS)

OS and DDFS will be analysed at the time of the IDFS analysis as per the multiple testing procedure (MTP) outlined in Section 4.2.6 and will use the same methodology and model as described above for the primary analysis of IDFS. The same pooling strategy as defined above for the IDFS end-point will be applied separately to the OS and DDFS end-points. Unadjusted analyses will also be done as a sensitivity analysis for OS and DDFS.

If applicable, a sensitivity analysis will be performed for DDFS and OS using the same model as described above for IDFS but based on all randomised patients confirmed to have *gBRCA* mutations by the central test. This analysis is only required if the analysis population differs from the primary ITT population (i.e. if any randomised patient is not confirmed to have a *gBRCA* mutation by the central test).

If the results of ER and PgR status from the local and central labs differ in >5% of randomised patients, then the stratified log-rank analysis will be performed for DDFS and OS using the central lab result to determine the HR status stratification factor and compared with the main OS/DDFS analysis result.

Subgroup analyses will also be conducted for DDFS and OS based on the same subgroups described above for IDFS. DDFS and OS will be analysed at the time of the primary analysis for IDFS.

The final OS analysis will be conducted once the trial follow up is complete (i.e. 15 years from first patient randomised assuming recruitment of 5 years).

In addition another analysis will be performed half way between the primary IDFS analysis and the final overall survival analysis (estimated around 10 years from first patient randomised but timings will be driven by the primary IDFS analysis once known). At this time point both DDFS and OS will be analysed and some alpha will be reserved for formal hypothesis testing. IDFS may also be updated if more information is available but this would be considered a supportive update of the primary analysis and no alpha will be reserved for IDFS.

For details on alpha spend and how this will be allocated across the planned analyses see Section 5

# 4.2.9 Contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, primary fallopian tube cancer and new primary peritoneal cancer

The incidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer will each be considered separately and be defined as the number and percentage of patients with documented evidence of contralateral invasive breast cancer, contralateral non-invasive breast cancer (contralateral DCIS), new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer regardless of when this occurs (i.e. does not need to be their first recurrence event).

The incidence of new contralateral breast cancer (invasive and non-invasive), new primary ovarian cancer, new fallopian tube cancer and new primary peritoneal cancer will be presented by randomised treatment group for the ITT population.

In addition, a table summarising all reported new cancers (i.e. not just breast, ovarian, fallopian tube or peritoneal cancers) will also be produced.

As described in Section 3.1.4, patients who have had a bilateral mastectomy prior to randomisation will be excluded from the analysis of new contralateral breast cancers (invasive and non-invasive) and patients who have had both ovaries removed prior to randomisation will be excluded from the analysis of new ovarian cancers and patients who have had their fallopian tubes removed prior to randomisation will be excluded from the analysis of new fallopian tube cancers. Males will be excluded from analyses of new primary ovarian, new primary fallopian and new primary peritoneal cancers.

The cumulative incidence of new primary contralateral invasive breast, new primary contralateral non-invasive invasive breast, new primary ovarian cancer, new primary fallopian tube cancer and new primary peritoneal cancer will be compared between treatment groups using competing risk analysis (Gray test, Fine and Gray 1999). Death will be considered a competing risk for each endpoint. In addition, bilateral mastectomy after randomisation will

be a competing risk for the contralateral breast cancer analyses, and bilateral oophorectomy after randomisation will be a competing risk for the new primary ovarian cancers analysis and removal of the fallopian tubes will be a competing risk for the new primary fallopian tube cancer analysis. Hazard ratios and 95% confidence intervals from competing risks regression analyses (Fine and Gray 1999) adjusted for randomised treatment group and the stratification factors will also be presented.

The same pooling strategy as defined above for IDFS, OS and DDFS end-points will be applied separately to each of new cancers endpoints. Unadjusted analyses will also be done as a sensitivity analysis for new cancers end points.

The Gray test and Fine and Gray models, not previously implemented in SAS, are now implemented in version 9.4.

- The data derivation requirements are similar to those of a traditional survival analysis, with "survival time" calculated as the time from randomisation to the occurrence of an event (or, here one of two or more possible events) or censored at the time of analysis if the event has not yet occurred. The key difference is a status variable which labels distinct codes for different causes of failure and a distinct code for censored observations.
- Cumulative incidence estimates will be plotted by treatment arm, for both the cause of interest and the competing risk(s). CI estimates are generated using the ODS option CIFPLOT in SAS 9.4.
- Proportional hazards model for the subdistribution of the competing risk, Fine and Gray models, will include the treatment arm and stratification factors and will be fitted using the '/ eventcode = #' option in the model statement of PHREG function in SAS9.4 to represent the event of interest (i.e. the new primary).
- The model will be stratified according to the pooling strategy.
- As with the proportional hazards model, tests will be performed to assess whether the Fine and Gray model is actually a reasonable fit to the data.
- The competing risk cumulative estimates will be presented for the 1<sup>st</sup>, 2<sup>nd</sup> and 3<sup>rd</sup> percentiles. The CIF estimates are generated using the OUTCIF option.

# 4.2.10 Analysis of patient reported outcomes

# **PRO** consent

In the US patients must consent specifically to collection of PRO data, the main study agreement is considered PRO consent for RoW.

# 4.2.10.1 Hypotheses and objectives

The hypotheses and measurement strategy focus on the fact that patients in the trial will be starting with significant decrements in HRQoL and high rates of symptoms at study entry (baseline) due to previous chemotherapy and local treatments (surgery with or without

radiation therapy). Therefore, the following hypotheses are proposed based on the expected toxicities of olaparib.

### **Primary PRO hypothesis**

Patients receiving olaparib may experience greater fatigue severity during treatment than those receiving placebo as measured by the FACIT-Fatigue scale at 6 and 12 months after randomisation.

# **Secondary PRO hypotheses**

- Patients receiving olaparib may experience greater GI symptoms (nausea/vomiting, diarrhoea and pain) severity during treatment than those receiving placebo as measured at 6 and 12 months after randomisation but no difference expected by 24 months after randomisation.
- There will be no difference in fatigue post discontinuation of study treatment as measured at 18 and 24 months.
- There will be no difference in QOL between the two treatment arms as measured by the global health status/QOL score and other functional sub-scales from the EORTC QLQ-C30 at 6, 12, 18 and 24 months after randomisation and patients will demonstrate improvements in functioning over time.

# **Primary PRO objective**

To determine the effect of olaparib on patient-reported fatigue at 6 and 12 months after randomisation as measured by the FACIT-Fatigue symptoms questionnaire.

# **Secondary PRO objectives**

- To determine the effect of olaparib on patient-reported GI symptoms (nausea, vomiting and diarrhoea) over time at 6, 12, 18 and 24 months as measured by the EORTC QLQ-C30 scale.
- To determine the effect of olaparib on patient reported fatigue over time at 6, 12, 18 and 24 months as measured by the FACIT-Fatigue questionnaire.
- To determine if there will be a difference in QOL between the two treatment groups over time as measured by the 2 item global health status/QOL score of the EORTC QLQ-C30 scale at 6, 12, 18 and 24 months and assess if patients demonstrate improvement in scores over time.
- To examine and compare the effect of olaparib over time on different functional sub scale scores as measured by the EORTC QLQ-C30 and assess if patients demonstrate improvement in functioning over time, with particular interest in the physical and emotional sub scales.

# 4.2.10.2 Administration of patient-completed questionnaire

### Time points for administration

The QOL questionnaires will be administered at the following time points:

- Baseline: Prior to randomisation after the consent form has been signed and eligibility confirmed.
- Following randomisation at 6 months, 12 months, 18 months and 24 months.

#### Administration instructions

After baseline, the QoL form will be administered at follow-up visits, so that when a follow-up visit is delayed, completion of the questionnaire may also be delayed. Patients who experience disease recurrence or diagnosis of a second primary cancer will not be expected to continue with the PRO assessments. Patients who discontinue study drug for other reasons will be expected to continue the PRO assessments per protocol schedule. Patients who never initiate study medication should not continue to complete PRO assessments. If a patient declines to complete a scheduled PRO assessment or if the questionnaire is not completed for any other reason (and cannot be completed by phone or mail), a Quality of Life Missing Data form should be submitted by the institution instead.

### 4.2.10.3 Statistical considerations for patient reported outcomes

# Statistical analyses

# Primary PRO endpoint - Fatigue

For the primary hypothesis, the composite fatigue score (FACIT-Fatigue questionnaire) measured at 6 and 12 months after randomisation will be compared between the two treatment arms using a mixed model for repeated measures analysis (MMRM) with adjustment for the corresponding baseline measurement. Separate analyses will be done for patients who have received prior neoadjuvant chemotherapy and patients who have received standard post-surgical adjuvant chemotherapy. Separate analyses are preferable because the timing of chemotherapy is expected to impact the fatigue outcome directly. Each comparison will be performed at the significance level of 0.05. No multiple comparisons adjustment will be employed since these outcomes evaluate the toxicity of the study treatment.

To further assess the effect of olaparib on fatigue over time (study treatment period and the year following) the composite fatigue score (FACIT-Fatigue questionnaire) measured at 6, 12, 18 and 24 months after randomisation will be compared between the two treatment arms using a mixed model for repeated measures (MMRM) analysis of all of the post baseline scores. Separate MMRM analyses will be done for patients who have received prior neoadjuvant chemotherapy and patients who have received standard post-surgical adjuvant chemotherapy. Further subgroup analysis by geographical region will be done if there are treatment differences at the higher level.

The model response variable will be average change from baseline and will include factors for treatment, visit and treatment by visit interaction, as well as covariates for baseline score and the baseline score by visit interaction. The treatment by visit interaction will remain in the model regardless of significance. Restricted maximum likelihood (REML) estimation will be used. The adjusted mean change from baseline estimates for each treatment arm, difference in the adjusted mean change from baseline estimates between the arms and corresponding confidence intervals will be presented by time point. Plots of the adjusted means changes (and corresponding confidence intervals) over time will also be presented.

An unstructured covariance matrix will be used to model the within-subject error and the Kenward-Roger approximation will be used to estimate the degrees of freedom.

If the fit of the unstructured covariance structure fails to converge, the following covariance structures will be tried in order until convergence is reached: toeplitz with heterogeneity, autoregressive with heterogeneity, toeplitz, and autoregressive.

Because this trial is being conducted internationally, responses to patient reported outcomes may be influenced by differences between country/language categories

Therefore, a subgroup MMRM analysis will be conducted for fatigue to assess consistency of treatment effect across geographic region (same categories as specified in Section 0). Separate MMRM analyses will be done for patients who have received prior neoadjuvant chemotherapy and patients who have received standard post-surgical adjuvant chemotherapy.

Adjustment for previous treatment exposures may also be considered as part of the secondary analyses. The following may be considered (by adding as a factor to the MMRM detailed above); previous radiation (yes vs. no), type of previous chemotherapy (anthracycline vs. taxane vs. both), previous platinum therapy (yes vs. no) and type of surgery (breast conserving vs. mastectomy).

As part of the secondary analyses, presence of treatment by hormone receptor status interaction will be investigated. Separate analyses will be performed for patients who have received prior neoadjuvant chemotherapy and patients who have received adjuvant chemotherapy. Each comparison will be performed at the significance level of 0.05. If the test is found to be statistically significant, the results of the treatment comparison will be presented by hormone receptor status

### **Secondary PRO endpoints**

A secondary analysis based on GI symptoms (nausea/ vomiting, diarrhoea and pain) from the EORTC QLQ-C30 symptom scale will be performed using the same MMRM model described above. Separate analyses will be done for patients who have received prior neoadjuvant chemotherapy and patients who have received standard post-surgical adjuvant chemotherapy.

The adjusted mean change from baseline estimates for each treatment arm, difference in the adjusted mean change from baseline estimates between the arms and corresponding

confidence intervals will be presented by visit. Plots of the adjusted means changes (and corresponding confidence intervals) over time will also be presented for nausea, vomiting and diarrhoea.

To assess if there are any difference in HRQoL, the 2 item global health status/QOL score assessed by EORTC QLQ-30 measured at 6, 12, 18 and 24 months after randomisation will be compared between the two treatment arms using the same MMRM model described above. Separate analyses will be done for patients who have received prior neoadjuvant chemotherapy and patients who have received standard post-surgical adjuvant chemotherapy. Plots of the adjusted means changes (and corresponding confidence intervals) over time will also be produced for the global health status/QOL score.

In addition, the 5 multi-item functional scales of the EORTC QLQ-C30 will be analysed using the MMRM model described above with particular interest in the emotional and physical subscales. Plots of the adjusted means changes (and corresponding confidence intervals) over time will also be produced.

All secondary analyses are considered exploratory and therefore no adjustments for multiplicity will be made. For each comparison, p-values (along with CIs) will be generated to help aid interpretation of the results using a nominal significance level of 0.05 (2-sided).

# Sample size consideration for PRO endpoints

We assume that half of triple negative patients and a quarter of hormone receptor positive patients will have received neoadjuvant chemotherapy and we anticipate that 95% of patients enrolled in the trial will complete the HRQoL instrument. In addition, adjusting downward to allow for 20% of missing data at the 12 months assessment point, we expect that data from 633 neoadjuvant and 735 adjuvant patients will be available (assuming that 15% of the total 1800 enrolled patients are ER and/or PgR positive/HER2 negative). These will be sufficient to provide statistical power of 93% and 96% correspondingly to detect a difference of 3 points on the FACIT-Fatigue scale score between treatment groups assuming a standard deviation of 10.9 (Cella et al 2002) (estimated SD of mean baseline score) and controlling  $\alpha$ -level at 0.05. A collection of PROs and QOL from all patients enrolled in the main trial will give us sufficient statistical power to detect important differences between the two treatment groups.

### Missing PRO data

If data for individual items are missing, imputation will be done according to the following: if less than 50% of the subscale items were missing (e.g. at most 2 of 5 items), the subscale score based on the non-missing items will be divided by the number of non-missing items and multiplied by the total number of items on the subscale. If at least 50% of the items are missing, that subscale will be treated as missing (not evaluable). If the scale is a single-item measure, a missing value will automatically be defined as 'Non-Evaluable'.

A certain amount of missing data is expected. The information from patients with missing data will be reviewed in order to determine whether data analytic procedures are likely to be

biased. Patients with missing data will be reviewed for imbalances in factors such as trial arm, treatment adherence, institution, and reason for non-adherence. When QOL data are missing at a particular time point, data from prior time points will be reviewed in order to investigate whether missing status was preceded by a significant change in QOL scores. In addition, we will investigate whether missing item status is related to other scores on the same questionnaire.

If there is no evidence from this review for dependence of the missingness mechanism on covariates or prior QoL scores, the data will be analysed assuming the data are missing at random (MAR).

If, on the other hand, the MAR assumption appears implausible, we will undertake to develop an appropriate analytic strategy to control for the potential bias and, if possible, to impute the missing values taking account of apparent dependencies in the data, for example by multiple imputation by chained equations. We will also present sensitivity analyses based on varying assumptions about the missing-data mechanism.

# 4.2.11 Pharmacokinetic analysis

The sample bioanalysis will be performed by and will be the responsibility of the clinical pharmacology scientist at AstraZeneca. The creation of a dataset suitable for non-linear mixed effects modelling (NONMEM) will be the responsibility of the AstraZeneca programmer and pharmacometrician. The NONMEM analysis will be the responsibility of the pharmacometrician and clinical pharmacology scientist at AstraZeneca. The plasma concentration summary and data listings will be the responsibility of Frontier Science.

A modelling analysis plan (MAP) will describe the population PK modelling objectives and approach. The plasma concentration-time data will be analysed (by NONMEM) in order to evaluate the pharmacokinetic characteristics of olaparib, quantify variability in the PK, identify demographic or pathophysiological covariates, which may explain the observed variability and explore exposure-response relationships to be reported outside of the CSR.

The olaparib plasma concentration data obtained from the samples collected in this study will be summarised and listed for the CSR but these data may be pooled with data from other studies in order to perform a population PK analysis. The PK/pharmacodynamic modelling methodology, results and conclusions will be reported in a separate PK/pharmacodynamic modelling report.

All plasma concentration data received will be presented in data listings based on the Full Analysis Set. A plasma concentration summary of the five samples taken on visit 4, Day 29 will be presented for patients in the PK analysis set, as defined in Section 2.1. Data from patients excluded from the PK analysis set and the reasons for exclusion from the PK analysis will be included in the data listings, but not in the summary. Extra measurements (such as unscheduled or repeat assessments) will also be excluded from the summary table but will be included in patient listings.

Plasma concentration data will be summarised using descriptive statistics, including n, arithmetic mean, standard deviation, coefficient of variation (%CV), median, minimum, and maximum values. Additionally, geometric means and geometric %CV (%GCV) will be reported. The geometric mean will be calculated as the exponential of the arithmetic mean calculated from data on a log scale. The %GCV will be calculated as " $100\sqrt{(\exp(s^2))}$  -1" where 's' is the standard deviation of the concentration data on a log scale.

For all data, descriptive statistics except for %CV and %GCV will follow the rounding convention of the individual data. Coefficients of variation (%CV and %GCV) will be reported to 1 decimal place. The concentration data will be reported to the same precision as the source data.

For descriptive statistics of concentrations, non-quantifiable (NQ) values of plasma concentrations will be handled as follows:

- If 50% or less of the plasma concentrations are NQ, the mean, standard deviation, geometric mean, %CV, and %GCV will be calculated by substituting the limit of quantification (LOQ) 0.0005 μg/mL for values which are NQ.
- If more than 50%, but not all, of the concentrations are NQ, the mean, geometric mean, standard deviation, %CV, and %GCV will be reported as not calculable (NC).

If all the concentrations are NQ, the geometric mean and mean will be reported as NQ and the standard deviation, %CV, and %GCV as NC.

### 4.2.11.1 PK level deviations

PK level deviations will be descried in more detail in the RAP. The following are considered deviations;

- Patient vomits on the PK sampling date or 3 days preceding the sampling date.
- Patient missed a dose or is on a reduced olaparib dose on the PK sampling day or the 3 days preceding the PK sampling day.
- Patient has taken a strong or moderate CYP3A inhibitor or inducer on any day prior to or on the day of PK sampling.
- PK samples incorrectly processed or analysed outside stability window
- PK sample was taken at a time which was significantly different from the protocol scheduled time.





### **4.2.13** Safety

Safety data will be summarised and listed only. No formal statistical analyses will be performed on the safety data. All safety data will be summarised by actual treatment group (olaparib or placebo). Any patient who received **at least one dose** of olaparib will be included in the olaparib group, even if the patient was randomised to receive placebo. However, some listings such as AEs listings will display the actual dose the patient received at onset of an AE.

### Adverse events

All AEs, both in terms of Medical Dictionary for Regulatory Activities (MedDRA) preferred term and common toxicity criteria for adverse events (CTCAE) grade, will be listed and summarised descriptively by count (n) and percentage (%) for each treatment arm. MedDRA dictionary will be used for coding and summaries will show the system organ class and preferred terms. Any AE occurring before olaparib/placebo treatment (i.e. before study day 1), and not worsening after study day 1 will be reported in the medical history table. These will be referred to as 'pre-treatment'.

The summary tables will include all AEs that occurred after the start of treatment up until the end of the 30 day follow-up period, referred to as "treatment emergent AEs", and those that start prior to treatment and then worsen following study day 1. The 30 day follow-up period will be defined as 30 days following discontinuation of olaparib/placebo treatment.

All reported AEs will be listed along with the date of onset, date of resolution (if AE is resolved), investigator's assessment of severity and relationship to study drug. Frequencies and percentages of patients reporting each preferred term will be presented (i.e. multiple events per patient will not be accounted for apart from on the episode level summaries).

Summary information (the number and percent of patients by treatment) will be tabulated for:

- All AEs
- All AEs causally related to study medication
- AEs with CTCAE grade 3 or higher
- AEs with CTCAE grade 3 or higher, causally related to study medication
- AEs with outcome of death
- AEs with outcome of death causally related to study medication
- All serious adverse events (SAEs)
- All SAEs causally related to study medication
- AEs leading to permanent discontinuation of olaparib/placebo

- AEs leading to permanent discontinuation of olaparib, causally related to olaparib/placebo
- SAEs leading to permanent discontinuation
- AEs leading to dose reductions
- AEs leading to dose interruptions
- AEs leading to dose reductions and interruptions
- AEs of special interest

An overall summary of the number and percentage of patients in each category will be presented, as will an overall summary of the number of episodes in each category. In addition, a truncated adverse event table of most common AEs, showing all events that occur in at least 5% of patients in any treatment arm will be summarised by preferred term, by decreasing frequency. This cut-off may be modified after review of the data.

Each AE event rate (per 1000 patient years) will also be summarised by preferred term within each system organ class. For each preferred term, the event rate will be presented and will be defined as the number of patients with that AE divided by the sum of the duration of therapy (for patients without the event) and the time to the AE (for patients with the event) in each group multiplied by 1000.

AEs will be assigned CTCAE grades (National cancer institute (NCI) CTCAE version 4.0) and summaries of the number and percentage of patients will be provided by maximum reported CTCAE grade, system organ class, preferred term and actual treatment group. Fluctuations observed in CTCAE grades during study will be listed.

In addition, adverse events with outcome of death, serious adverse events, adverse events leading to discontinuation of treatment and adverse events causally related to olaparib/placebo will be listed.

A summary of deaths will be provided with number and percentage of patients by actual treatment group, categorised as:

- Primary cause of death
- Time to death from last dose
  - <=30 days
  - >30 days

A corresponding listing will also be produced.

# **Summary of long-term tolerability**

To assess long-term tolerability, provided that there are a sufficient number of patients with events to warrant it, prevalence plots, life table plots and cumulative incidence plots will be presented for each of nausea, vomiting, anaemia, neutropenia, thrombocytopenia, and fatigue and asthenia, provided there are  $\geq 10$  events, see table below for preferred terms to identify the AE.

Table 8 AEs for summary of long term tolerability

| AE | Preferred terms |
|---|---|
| Nausea | Nausea |
| Vomiting | Vomiting |
| Anaemia | Anaemia, Haemoglobin decreased, Haematocrit decreased, Red<br>blood cell count decreased, Erythropenia, Anaemia macrocytic,<br>Normochromic anaemia, Normochromic normocytic anaemia,<br>Normocytic anaemia |
| Neutropenia | Febrile neutropenia, Granulocyte count decreased,<br>Granulocytopenia, Neutropenia, Neutropenic infection, Neutropenic<br>sepsis, Neutrophil count decreased, Idiopathic neutropenia,<br>Agranulocytosis |
| Thrombocytopenia | Platelet count decreased, Platelet production decreased,<br>Thrombocytopenia, Plateletcrit decreased |
| Fatigue & asthenia | fatigue and asthenia |

A prevalence plot provides information on the extent to which the events may be an ongoing burden to patients. The prevalence at time *t* after first dose of study treatment is calculated as the number of patients experiencing the event divided by the number of patients receiving study treatment or in safety follow-up at time *t*; generally, *t* is categorised by each day after dosing. The prevalence is plotted over time split by treatment arm. Multiple occurrences of the same event are considered for each patient but a patient is only counted in the numerator whilst they are experiencing one of the occurrences of the event.

For each AE, median time to first onset of the AE will be presented in patients in the Safety Analysis Set by actual treatment group. Patients who did not experience the AE will be censored at the end of their safety follow-up. Summary tables of time to first onset for each AE will also be produced (e.g. 1-28 days, 29-56 days, 57-84 days, 85-112 days, >112 days). Median duration of the AE will be presented in patients who experienced each AE.

Median time to first occurrence is calculated using Kaplan-Meier. Patients who do not experience the event are censored at the end of the survival at either the end of safety follow-up or at data cut-off if they are still in follow-up at data cut-off. The ODS options 'Quartiles' from PROC LIFETEST can be used to identify the median time to first occurrence.

Duration of first adverse event is defined as end date - start date + 1. If there is no end date recorded then the end of safety follow-up or (if they are still in follow-up) the data cut-off will

replace the end date. The median duration will be calculated including the first occurrence of the AE per patient across all the patients that experience the adverse event.

Number of patients with a first event that has a resolution is the count of the patients with first event where the adverse event outcome = 'Resolved'.

Summary statistics for time to first occurrence are calculated only for patients who experience the adverse event, summary statistics include; n, mean, median, min, and max.

A life table plot will be used to describe the time to onset of the event and specifically when patients are at most risk of first experiencing the event. The hazard, or in other words, the probability of having an AE in a specified time period (e.g. 0-1 months, 1-3 months, 3-6 months, etc.) given that the patient reaches that time period without having an event will be plotted for each time period split by treatment.

A cumulative incidence plot, which is a plot of the raw cumulative incidence and cumulative incidence function over time, will be produced with the treatment arms presented on separate plots. The raw cumulative incidence will be the actual probability that a patient will have experienced their first occurrence of the event by a given time point. The cumulative incidence function will estimate the cumulative incidence if the data cut-off had not been imposed and all patients had completed safety follow-up. The raw cumulative incidence is derived by calculating the number of subject events occurring up to a given month, divided by the number of patients still taking study medication at that month.

A summary of AESI occurring > 30days post treatment will also be included.

### Laboratory assessments

Box-plots of absolute values and change from baseline for continuous laboratory assessments will be presented, with AZ project defined reference ranges indicated. For all continuous key laboratory parameter assessments, absolute value, change from baseline and percentage change from baseline will be summarised using descriptive statistics at each scheduled assessment time by actual treatment group. For categorical laboratory assessments, shift from baseline will be summarised using frequency and proportion at each scheduled assessment time by actual treatment group.

Shift tables for laboratory values by worst common toxicity criteria (CTC) grade will be produced, and for specific parameters separate shift tables indicating hyper- and hypodirectionality of change will be created. For parameters with no CTCAE grading, shift tables from baseline to worst value on-treatment will be provided (i.e. on-treatment is defined as data collected up until the last dose of olaparib/placebo). Shift tables for appropriate urinalysis values by worst grade may be also provided as appropriate.

# Summary of Hy's law

**Hy's law**: Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)  $\geq 3x$  Upper Limit of Normal (ULN) together with Total Bilirubin (TBL)  $\geq 2x$ ULN.

**Potential Hy's law**: AST or ALT  $\ge 3x$  ULN together with TBL  $\ge 2x$ ULN at any point during the study following the start of study medication irrespective of an increase in Alkaline Phosphatase (ALP).

For Hy's law and Potential Hy's law the elevation in transaminases must precede or be coincident with (i.e. on the same day) the elevation in TBL, but there is no specified timeframe within which the elevations in transaminases and TBL must occur.

Maximum on treatment ALT and AST by maximum total bilirubin for assessing Hy's Law criteria will be summarised.

An eDISH plot of maximum alanine aminotransferase (ALT) versus maximum total bilirubin, both expressed as multiples of upper limit of normal (ULN), will be produced. The eDISH plot will be repeated for maximum aspartate aminotransferase (AST) versus maximum total bilirubin.

Liver biochemistry test results over time for patients meeting Potential Hy's law criteria with elevated ALT or AST, and elevated total bilirubin (at any time) will be plotted.

Individual subject data will be presented for subjects with potential Hy's Law.

Clinically significant laboratory results will be flagged and listed. Reference ranges will also be listed. All laboratory summaries and listings will be presented by actual treatment group.

### Vital signs

Box plots for absolute values and change from baseline in systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate and body temperature will be produced. Vital signs (SBP, DBP, heart rate and body temperature) will be summarised over time in terms of absolute values and changes from baseline at each scheduled measurement by actual treatment group. Height, weight and vital signs data at baseline will be summarised in baseline characteristics summaries by planned treatment group.

### **ECGs**

Overall evaluation of ECG at baseline will be summarised by planned treatment. The results will be classified as normal or abnormal with abnormal having sub-categories of "clinically significant" and "not clinically significant". Any clinically significant ECG assessments on whilst on study treatment will be listed.

## 4.2.14 Treatment exposure

The following summaries related to study treatment will be produced for the Safety Analysis Set by treatment received:

- Total intended exposure of olaparib/placebo.
- Actual exposure of olaparib/placebo.

- Number of days on 300 mg olaparib/placebo bd. = actual exposure for the dose assigned.
- Reasons for dose reductions, dose interruptions, and dose reduction & interruption of olaparib/placebo. Dose reductions and dose interruptions will be based on investigator initiated dosing decisions. Dose interruptions/reductions due to "Subject non-compliance" will be omitted from these summaries.
- Number of dose interruptions of olaparib/placebo that last for a period of three days or more.
- PID and RDI of olaparib/placebo (entire intended treatment period).

### 4.2.15 Imputation for Missing/Partial Dates

Data management will query all missing or partial fields in the eCRF, however it is expected that some queries will not be resolved. To limit the impact on the analyses and reporting, some imputations will be applied if dates relating to adverse events, concomitant medication or efficacy events are partial or missing (see Table 9 below). For AE and concomitant medications, imputation methods will be used on partially missing or wholly missing start or end dates to decide if an observation is treatment emergent.

Imputed dates will not be displayed in listings and duration of AE/Medication will not be calculated for imputed dates. The partial date imputation will follow ADaM conventions which populates the numeric date variables with the imputed date and adds a flag variable to the dataset that indicates the level of imputation.

 Table 9
 Imputation for missing or partial dates

| Field | Missing element(s) | Rule |
|---|---|---|
| Start Date for Any AE/Concomitant Medication | Any | Ensure that the new imputed date is not after the end date* of the AE or Medication or after the data cut-off date. |
| | | *provided there is more information known. |
| | Day | If month and year same as month and year of first dose of study drug then impute first dose date, else impute first day of the month |
| | Day and month | If year same as year of first dose of study drug then impute first dose date, else impute 1st January |
| | Day, month and year | Impute first dose date unless it is after the end date in which case impute the 1 <sup>st</sup> January of the same year as the end date |
| Date 12th June 2019 | | |
|---|---|---|
| End Date for AE/Concomitant Medication | Any | Ensure that the new imputed date is not before the start date (including imputed start date) of the AE or Medication or after the data cut-off date. |
| | Day | If month and year same as month and year of last dose of study drug then impute last dose date, else impute the last day of the month |
| | Day and month | If year same as year of last dose date then impute last dose date, else impute 31st December |
| | Day, month<br>and year | Check if AE/Medication is still ongoing and when it started in relation to study drug. (1) If ongoing flag is missing, assume AE/Medication is still being taken and do not impute, (2) If AE/Medication has stopped and start date is prior to first dose date then impute first dose date (3) If AE/Medication has stopped and start date is on or after first dose date then impute last dose date |
| Date of death | Day | If month and year same as month and year of date of last contact (see Section 3.1.2), then impute date of last contact, else impute first day of the month. |
| | Day and month | No imputation |
| | Day, month and year | No imputation |
| Recurrences and second primary malignancies | Day | If month and year same as month and year of date of last disease evaluation (see Section 3.1.1), then impute date of last disease evaluation, else impute first day of the month. |
| | Day and month | No imputation |
| | Day, month and year | No imputation |

## 4.2.16 Central pathology result timepoint for analysis

Central pathology review samples are analysed by IEO, the results from these samples are used in the summary of patients' central receptor status (ER, PgR and HER2) and in central pathology review sensitivity analysis which is triggered by the difference between local and central HR status.

Adjuvant patients are expected to have an archival tumour sample, neoadjuvant patients can have both archival and post neoadjuvant, however both are not compulsory (as of protocol version 2), thus resulting in some patients having central pathology review results for more than one timepoint. For the purpose of the CSR analysis specified in the SAP it is key to have a single central pathology review result for ER, PgR and HER2.

The following process was agreed by the study team (reference memorandum) for identifying the single central pathology review result to be used in the summary tables and in the sensitivity analysis using the central pathology results.

- When a patient has central pathology review results for more than one timepoint, sites were asked which sample was used to determine eligibility. If sites can confirm which of the archival or surgical sample was used then this is used as the central pathology result.
- In the case that the site cannot provide an answer the earliest sample date will be used to identify which result should be used for the analyses.

The scenario could also occur where more than one specimen is taken at a single time point, resulting in a single accession number and more than one sample result.

- If the samples provide the same result for HR and HER2 then the central pathology result will be the combined result.
- If the central result samples are not the same then accession number and sample that has the same HR result as the eCRF will be identified and used as the central result.

Appendix E contains the specification for identification of a patients central pathology review result.

# 5. INTERIM ANALYSES

A superiority interim analysis of IDFS will occur when half the events required for the final analysis (165 events) have been observed in the first 900 patients (50% of the planned total recruitment). This provides a cohort of patients with a similar level of maturity that is planned for the final analysis. The interim analysis is predicted to be October 2019 (80% confidence interval: March 2019 - August 2020).

If the interim analysis is triggered then all analyses, with the exception of the exploratory analyses will be generated.

The same pooling strategy as defined above (section 4.2.7.1) for the primary analyses will be applied at the interim. Two populations will be analysed at the interim analysis based on the analysis methods described in Section 4.2 for IDFS:

- 1 Primary: ITT population (all patients randomised, estimated 254 events (80% confidence interval: 226 289).
- 2 Supportive: Mature cohort population (first 900 patients randomised, 165 events anticipated).

The inclusion of a mature cohort population at the interim provides confidence that any observed treatment effect from the interim ITT population is maintained with longer-term follow up. It is anticipated, based on the data available at the time of the protocol amendment (version 5) and on the assumed recruitment and event rate, that the interim analysis will occur approx. 5.3 years after the first patient is randomised and that all patients will have been randomised. The mean follow-up is expected to be 27 months in the ITT set, and 34 months in the mature cohort.

Evidence of superiority for IDFS would only be determined at the interim if the results from both analysis populations provide evidence of a sustainable clinically relevant treatment effect. More specifically, the result in the ITT population would need to have met the statistical threshold defined below. When the statistical threshold is met in the ITT population, the result in the mature cohort (i.e. HR) would need to be of a similar magnitude, such that the IDMC would consider it supportive of the ITT result. This will have added confidence in the result in the ITT population. Statistical significance is not required for the mature cohort population. This analysis will be regarded as supportive, based on a cohort of patients with longer term follow up. This to aid interpretation of the result in the ITT population based on interim data. Other outcome measures such as 3 year IDFS rate will also be presented to aid the interpretation of the HRs (particularly in the case where the assumption of proportional hazards may not hold). KM plots will also be produced for IDFS.

The test mass alpha for IDFS (1 sided 2.5%) will be split between the final and the interim analysis using a bespoke spending function where a fixed significance level will be assigned at the interim and the remaining significance level assigned to the final analysis, taking account of correlation (Stone 2009). A 2-sided significance level of 0.005 will be assigned to the interim analysis so that a highly significant and clinically relevant result will need to be observed to declare superiority on IDFS. As an illustration, if 70% of the total required 330 IDFS events have occurred in the ITT population at the interim then the observed HR would need to be <0.701 for superiority to be declared based on p<0.005 and the HR in the mature cohort would need to be supportive of the ITT result. The significance level for the final IDFS analysis would be 0.0493 in this example.

If the null hypothesis for IDFS is rejected at the interim for the ITT population then secondary endpoints (DDFS and OS) will be tested based on the MTP procedure outlined in Section 4.2.2 using the significance levels provided in Table 10. If IDFS is not significant at

the interim, DDFS and OS will not be tested at the IDFS interim and the significance level allocated to the IDFS interim for DDFS and OS will not be allocated to later time points.

Similar to IDFS, a bespoke spending function will be applied to the secondary endpoints OS and DDFS where a fixed significance level will be assigned to each analysis time point and the remaining significance level assigned to the final analysis time point controlling the overall type 1 error at the pre-specified alpha amount (Stone 2009). Provided the last analysis is known in advance of the penultimate one then the remaining alpha can be split to ensure that some alpha is always reserved for the final analysis. This approach allows flexibility in the number of analyses while appropriately controlling the overall type 1 error. Three analyses are planned for DDFS and four for OS for which some alpha will be reserved for significance testing. If additional analyses are required beyond the planned analyses and some alpha is still available for testing then any remaining alpha can be further split to strongly control the type 1 error (based on process described above). If no alpha remains then the additional analyses will be considered supportive updates of the already conducted analyses.

Given the split in alpha between DDFS and OS, if OS is significant based on the assigned significance level then the alpha assigned to OS will be recycled to DDFS and split across the planned analyses (and vice versa if DDFS is significant alpha for DDFS will be recycled to OS and split across analyses). The recycled alpha will be split based on the ratio of the originally assigned alpha split. For example if the original alpha allocation was split 1/3 for each analysis time point then the recycled alpha would also be split 1/3 across each analysis time point. For example, at the first interim analysis, assume IDFS is statistically significant and the secondary endpoint OS is also statistically significant. The significance level for testing DDFS is therefore  $0.005 + (\text{alpha assigned to OS recycled to DDFS and split across the planned analyses), i.e. <math>0.005 + (1\% * 0.005/0.04 = 0.00125) = 0.00625$ , or alternatively thought of as 0.005 \* 5/4.

Secondary endpoints will be assessed based on the ITT population. Table 10 shows the different 2-sided significance levels that will be applied to the primary and secondary endpoints across the planned analyses, as well as the total alpha spend for each endpoint. Note: the significance level for the final analyses of each endpoint will be calculated using the relevant correlation. This is based on the actual number of events for each analysis, the previous alpha spend and the total allocated alpha for that endpoint.

The significance level for the final analyses of each endpoint can be calculated using the software package EAST by selecting the 'boundary family p-value (HP)' option. The following information is required:

- Total allocated alpha for the endpoint being analysed
- Significance levels used for all previous analyses
- Proportion of events at each previous analysis (derived as actual number of events at analysis time point divided by total number of events at final analysis time point)

Edition Number 3.0 Date 12th June 2019

Table 10 Summary of 2-sided significance levels and total alpha spend across the endpoints and analyses

| Endpoints | Interim<br>analysis | Final IDFS analysis | DDFS and OS analysis | Final OS<br>analysis | |
|---|---|---|---|---|---|
| Estimated timings from | | | | | |
| FSI [1] | 5.3 years | 6.5 years | 10 years | 15 years | |
| | Significance level | Significance level | Significance<br>level | Significance level | Total alpha<br>spend (2-<br>sided) |
| IDFS | 0.005 | TBC [2] | N/A | N/A | 5% |
| If IDFS is statistically significant and alpha is not recycled between secondary endpoints at the analysis [3] | | | | | |
| DDFS | 0.005 | 0.02 | TBC* | N/A | 4% |
| OS | 0.002 | 0.003 | 0.004 | TBC* | 1% |
| If IDFS is statistically significant and alpha is recycled between secondary endpoints at the analysis [4] | | | | | |
| DDFS | 0.00625 | 0.025 | TBC* | N/A | 5% |
| OS | 0.01 | 0.015 | 0.02 | TBC* | 5% |

- [1] FSI: first subject randomised
- [2] TBC: to be calculated; significance level to be calculated once relevant correlation based on the actual number of events for each analysis is known taking account of previous alpha spend and total allocated alpha
- [3] i.e. both OS and DDFS rejected or accepted
- [4] If the null is rejected for OS and not for DDFS then alpha will be recycled to DDFS from OS. If the null is rejected for DDFS and not for OS then alpha will be recycled to OS from DDFS.

The IDMC will review the data from the interim analysis. The boundaries defined by the interim p-values for efficacy will be used as guidelines by the IDMC along with all other relevant trial information, including the safety data, to decide if it is appropriate to make a recommendation other than that to continue the trial as planned.

Simultaneously to the interim analysis for superiority, an assessment of futility will be performed. This futility assessment will be based on the probability of eventually showing statistical significance for the primary endpoint when the final number of IDFS events (n=330) is reached (Lachin 2005). The determination of this probability will be conditional on the observed data in the ITT population at the time of the interim analysis for superiority and on the assumed hazard ratio for the alternative hypothesis (IDFS HR=0.7). If the probability is less than 0.1, the IDMC will consider the option of declaring futility.

This study will use an IDMC whose members include therapeutic area experts and statisticians who are not employed by AstraZeneca and do not have any major conflict of interest. BIG,

AstraZeneca, CTEP and NSABP will jointly select members of the IDMC and the IDMC will report their recommendations to the steering committee.

The IDMC will meet approximately every 6 months and will review ongoing study progress including safety and, when appropriate, efficacy data. They will also review the data presented at the time of the protocol-defined interim analysis. The IDMC will have the ability to recommend suspension of enrolment if safety concerns are identified at any of the six monthly assessments. At the interim analysis, both efficacy and safety will be reviewed and trial recommendations will be based on the totality of the data. The IDMC can recommend changes to the trial, including stopping of the trial, if they have concerns over the benefit risk profile for olaparib.

Reports for the IDMC will be prepared by an Independent Statistical Centre (ISC) and will be presented to the IDMC in closed session. Following review of data, the IDMC will make a recommendation regarding the future conduct of the trial to the steering committee. The IDMC recommendation will not contain any unblinded information or any information related to treatment outcomes of the trial. A separate IDMC Charter will be developed defining the responsibilities and procedures for the IDMC.

# 6. CHANGES OF ANALYSIS FROM PROTOCOL

The analyses described here are based on the protocol edition 5, dated 18 May 2018, with file name "OlympiA Protocol v5 (Amendment) effective 18-May-2018.pdf".

# 6.1 Censoring of patients not at risk for disease evaluated

The protocol states the following with regards to censoring for IDFS, DDFS and OS

- Patients who have not had a recorded IDFS event at the time of the analysis will be censored at the date of their last disease evaluation.
- Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
- Patients who do not have documented evidence of DDFS at the time of the analysis of DDFS will be censored at the date of their last clinical examination (i.e. last physical exam or radiological evaluation).

The study team identified that patients had been randomised that are not at risk for the endpoint evaluated in OlympiA. The decision by the SST and wider AZ team was to censor these patients at 0.5 days (rationale for 0.5 days is discussed previously).

This process would leave the information in the database as submitted by the investigator unchanged and define the ITT population as all randomized patients.

We specify above that observations from patients who are retrospectively (after randomization) discovered to have had an IDFS event prior to randomization will be considered in the data analysis as censored 0.5 days this assures that the baseline number at

risk on the Kaplan-Meier curves matches the number in the ITT population reported in the CONSORT diagram).

This approach has been widely used for the analyses of adjuvant breast cancer trials by cooperative groups for decades, this approach does not require a protocol amendment, just a specification in the SAP about how data will be handled for the analysis. The 3 scenarios under which patients are censored at 0.5 days are:

- Patients who have had an event prior to randomisation.
- Patients who were identified as inadvertent randomisations (i.e. patient was randomised and the site noticed afterwards that they should not have been randomised, they have had no follow-up nor did they receive treatment).
- Patients who have withdrawn consent, received no treatment, and will not be providing any follow-up data.

#### 7. REFERENCES

#### Anderson et al 2004

Anderson P.K, Hansen, M.G., Klein, J.P. Regression analysis of restricted mean survival time based on Pseudo-observations. Lifetime Data Anal. 2004; 10(4): 335-350.

#### Bernhard et al 2007

Bernhard J, Zahrieh D, Castiglione-Gertsch M, et al. Adjuvant chemotherapy followed by goserelin compared with either modality alone: the impact on amenorrhea, hot flashes, and quality of life in premenopausal patients—the International Breast Cancer Study Group Trial VIII. J Clin Oncol 2007; 25:263-270.

#### Cella et al 2002

Cella D, Eton DT, Lai JS, et al. Combining anchor and distribution-based methods to derive minimal clinically important differences on the Functional Assessment of Cancer Therapy (FACT) anemia and fatigue scales. J Pain Symptom Manage 2002; 24(6):547-561

#### Collett 2003

Collett, D. (2003) Modeling Survival Data in Medical Research. 2nd Edition, Chapman @ Hall/CRS A CRC Press Company, London, New York, Washington, D.C.

#### Cortazar et al 2014

Cortazar P, Zhang L, Untch M, et al. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. *The Lancet*, 2014: 384(9938), pp.164-172.

#### Dent et al 2007

Dent R, Trudeau M, Pritchard K, Hanna W, Kahn H, Sawka C, Lickley L, Rawlinson E, Sun P, Narod S. Triple-Negative Breast Cancer: Clinical Features and Patterns of Recurrence. Clinical Cancer Research 2007; 13(15), 4429-4434.

## Dmitrenko et al 2005

Dmitrienko A, Molenberghs G, Chuang-Stein C, Offen W. 2005 Analysis of Clinical Trials Using SAS: A Practical Guide. Cary, NC. SAS Insitute Inc

#### Fine and Gray 1999

Fine, J. and Gray, R. A Proportional Hazards Model for the Subdistribution of a Competing Risk, Journal of the American Statistical Association, 1999: 94, 496–509.

#### Gail and Simon 1985

Gail M, Simon R. Testing for qualitative interactions between treatment effects and patient subsets. Biometrics 1985;41:361-72.

#### Glimm et al 2009

Glimm, E., Maurer, W., and Bretz, F. Hierarchical testing of multiple endpoints in group-sequential trials. Statistics in Medicine 2009;29, 219–228.

#### **Grambsch and Therneau 1994**

Grambsch P, and Therneau T. Proportional hazards tests and diagnostics based on weighted residuals. Biometrika 1994; 81: 515-26.

#### Hudis et al 2007

Hudis CA, William E, Barlow JP, Costantino RJ, Gray KI, Pritchard J-AW, et al. Proposal for Standardized Definitions for Efficacy End Points in Adjuvant Breast Cancer Trials: The STEEP System. J Clin Oncol 2007;25(15):2127-32.

# Jeruss et al 2008

Jeruss SJ, Mittendorf EA et al. Combined Use of Clinical and Pathologic Staging Variables to Define Outcomes for Breast Cancer Patients Treated With Neoadjuvant Therapy. J Clin Oncol 2008; J Clin Oncol 26:246-252.

#### Lachin 2005

Lachin, J. M. (2005). A review of methods for futility stopping based on conditional power. Statist. Med., 24: 2747–2764. Statist Med 24:2747-2764

#### Mittendorf et al 2011

Mittendorf EA, Jeruss JS, Tucker SL, Kolli A, Newman LA, Gonzalez-Angulo AM, Buchholz TA, Sahin AS, Cormier JN, Buzdar AU, Hortobagyi GN, Hunt KH. Validation of a Novel Staging System for Disease-Specific Survival in Patients With Breast Cancer Treated With Neoadjuvant Chemotherapy. Journal of Clinical Oncology 2011 vol 29 no 15 may.

Personal communication with B-38 protocol statistician, Joseph Costantino, 12/01/2015, Email.

#### Pintilie M.

Competing risks: A practical perspective. Wiley.

# **Robins and Tsiatis 1991**

Robins JM, Tsiatis AA. Correcting for noncompliance in randomized trials using rank preserving structural failure time models. Communications in Statistics - Theory and Methods 1991; 20:2609-2631.

#### **Stone 2009**

A Stone. The application of bespoke spending functions in group-sequential designs and the effect of delayed treatment switching in survival trials. Pharmaceutical statistics 2009; 9, 151-161

#### Swain et al 2013

Swain S, Tang G, Geyer C, Rastogi P, Atkins J, Donnellan P, Fehrenbacher L, Azar C, Robidoux A, Polikoff J, Brufsky A, Biggs D, Levine E, Zapas J, Provencher L, Northfelt D, Paik S, Costantino J, Mamounas E, Wolmark N. Definitive Results of a Phase III Adjuvant Trial Comparing Three Chemotherapy Regimens in Women With Operable, Node-Positive

Breast Cancer: The NSABP B-38 Trial. Journal of Clinical Oncology 2013; 31(26), 3197-3204

#### Therneau and Grambsch 2000

Therneau T and Grambsch P.Modeling Survival Data: Extending the Cox Model. Springer, New York. 2000; ISBN 0-387-98784-3.

#### Therneau 2015

Therneau T. A Package for Survival Analysis in S. version 2.38, 2015. https://CRAN.R-project.org/package=survival.

#### Yellen et al 1997

Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage 1997; 13(2), 63-74.

Clinicaltrials.gov, (2015). A Study of Palbociclib in Addition to Standard Endocrine Treatment in Hormone Receptor Positive Her2 Normal Patients With Residual Disease After Neoadjuvant Chemotherapy and Surgery - Full Text View - ClinicalTrials.gov. [online] Available at: https://clinicaltrials.gov/ct2/show/NCT01864746?term=PENELOPE&rank=2 [Accessed 9 Apr. 2015].

# 8. APPENDIX A

### **Background**

To support the addition of the ER+ cohort in protocol version 4 a simulation study was undertaken with the objective to predict accrual of events and therefore the timing of the interim and primary analyses.

The simulation study included relevant operating characteristics for the anticipated possible proportions enrolled in each of the 4 subgroups, survival was modelled by piecewise exponential distribution for which annualized hazard according to the respective subgroups were taken from the most recent published data (Dent et al 2007, Cortazar et al 2014, B 38 data, and GBG data).

Following the observation of lower than anticipated event rate, it was clear that the published data used for the simulations were too pessimistic with respect to event rates for the Triple negative BRCA carrier population that would be recruited into OlympiA since 2014.

Further predictions were run using the current data (extract date 10Nov2017) and applying AZ's 'Shiny' oncology event prediction R package. A survival model assuming a Weibull distribution was fitted to the previous study data and used to predict future survival times. Whilst the simulation study simulated over varying proportions enrolled in each sub group, by using the current data, the predictions were based on 1153 patients of whom 15% were ER+ and the ratio of Adjuvant to Neoadjuvant was roughly 1:1. An 8% drop-out rate for the first 12 months, not previously included, was incorporated based on the rate observed so far. The program predicted the future enrolment to 1800 based on the recent observed enrolment rate.

Given the predictions for timing of the interim and primary analysis it was decided to increase the sample size to 1800 and for the power to remain at 90%. Because the event rate was lower than anticipated rather than higher than anticipated, the restriction to have a minimum 2 year follow-up after the last patient enrolled could be removed. Patient enrolment would continue about one year longer than originally anticipated and more patients would be enrolled, thus providing an increase in the number of patient years of follow-up at the time of primary analysis even without the 2 year minimum follow-up criteria.

Date 12th June 2019

#### **APPENDIX B**

As described in Section 3.3.2, treatment exposure of olaparib/placebo will be defined as follows:

- Total (or intended) exposure = last dose date first dose date + 1
- Actual exposure = intended exposure total duration of dose interruptions, where intended exposure will be calculated as above.
- Number of days on 300 mg olaparib/placebo bd. = actual exposure for the dose assigned.

Example of patient who permanently discontinued during a dose Table 11 interruption, documented on eCRF page "Administration of Olaparib/Placebo"

| Start date | Stop date | Total daily dose (mg) | Was dose reduced? | Reason dose reduced | Was treatment interrupted? | Reason for interruption |
|---|---|---|---|---|---|---|
| 23/01/2015 | 14/02/2015 | 600 | No | | No | |
| 15/02/2015 | 28/02/2015 | 600 | No | | Yes | Adverse<br>Event |
| 02/03/2015 | 13/03/2015 | 500 | Yes | Adverse<br>Event | No | |
| 14/03/2015 | 15/03/2015 | 500 | No | | Yes | Adverse<br>Event |

When treatment stops (on 15/03/2015 in this example), the investigator will then complete the "Treatment completion" page of the eCRF. The stop date recorded on the administration page should correspond with the date of last dose on the completion page. In this example, the reason for non-completion (discontinuation of the study drug) should be recorded as adverse event, matching the reason for interruption.

However, there is an exception where reason for interruption can differ from reason for noncompletion. When a patient experiences an AE and interrupts treatment, the reason for interruption should be recorded as AE. If the patient does not restart treatment due to disease progression, resulting in discontinuation of treatment, the reason for non-completion should be recorded as progression of disease. Therefore, the reason of interruption does not match the reason of non-completion.

# 10. APPENDIX C

Figure 4 Examples of dose intensity for olaparib/placebo dosing



Patients 1-4 progressed on Day 15, so the intended dose through to progression was 14 \* 300 mg \* 2 of olaparib/placebo = 8400 mg.

All 4 patients received less treatment due to:

- Missed/forgotten doses (Patient 1)
- Dose reduction and early stopping (Patient 2)
- Dose interruption (Patient 3)
- Early stopping (Patient 4)

Patient 1: 
$$RDI = PID = ((12 * 300 \text{ mg} * 2) + (2 * 300 \text{ mg}))/8400 \text{ mg} = 93\%$$

Patient 2: RDI = 
$$((7 * 300 \text{ mg} * 2) + (4 * 150 \text{ mg} * 2))/(11 * 300 \text{ mg} * 2) \text{ mg} = 82\%$$
  
PID =  $((7 * 300 \text{ mg} * 2) + (4 * 150 \text{ mg} * 2))/(8400 \text{ mg} = 64\%)$ 

Patient 3: PID = 
$$(7 * 300 \text{ mg} * 2)/8400 \text{ mg} = 50\%$$
  
RDI =  $(7 * 300 \text{ mg} * 2)/4200 \text{ mg} = 100 \%$ 

Patient 4: RDI = 
$$((5 * 300 \text{ mg} * 2) + (1 * 300 \text{ mg}))/(6 * 300 \text{ mg} * 2) = 92\%$$
  
PID =  $((5 * 300 \text{ mg} * 2) + (1 * 300 \text{ mg}))/(8400 \text{ mg} = 39\%)$ 

Due to the eCRF design, the actual cumulative dose does not capture all missed or forgotten doses within an individual day. This will be recorded as if the patient took a full daily dose, which could lead to an overestimation of RDI and PID.

# 11. APPENDIX D

GailSimon macro (Dmitrenko et al 2005)



#### 12. APPENDIX E

Derivation of central pathology review result for analysis.

Central pathology review specification:

# 12.1 Purpose

The detail contained in this appendix aims to specify the process for identifying the central pathology review result for each patient, depending on what we receive from IEO.

The study team agreed the following;

- 1 If the site cannot identify which time point the patient was randomised under then the earliest should be used.
- If there are duplicate accession numbers for a time point that has been identified as the one randomised under then the following algorithm will be applied.
  - o If all the results are the same then the combined result is used
  - o If the results are not the same then the sample in which the HR status is the same as the HR status reported on the eCRF (i.e. the local result) is used.

See HR status memo (AZ document) for further details.

# 12.2 Derivation of Central pathology results from the data provided by IEO

Table 12 IEO data HR status (ER & PgR) and HER2 results (See DTS)

| Variable name | Variable label | Valid values |
|---|---|---|
| ER | % of estrogen receptor expression | 0-100,NA |
| PgR | % of progesterone receptor expression | 0-100,NA |
| HER2 IHC | HER2 score | 0,1,2,3,NA |
| HER2 IHC % | % of HER2 expression | 0-100,NA |
| HER2 FISH | HER2 Fish result | amplified, not amplified, NA |

Table 13 Derivations for classifications of HR status and HER2 results for CSR

| | Classification presented in the CSR | Derivation from IEO data |
|---|---|---|
| ER status | Positive, Negative, Missing | ER positive is defined as >=1% ER receptor expression |
| PgR status | Positive, Negative, Missing | PgR positive is defined as >=1% PgR receptor expression |
| HR status | Positive, Negative, Missing | HR positive is defined as >=1% ER or PgR receptor expression. |
| HER2 FISH results | Amplified, Not amplified, Not assessable,, Missing | Amplified = Amplified |
| | | Not amplified = Not amplified |
| | | NA = Not assessable |
| | | " = Missing |
| HER2 IHC results | 0, 1+ ,2+ , 3+, NA, Missing | 0 = 0 |
| | | 1 = 1+ |
| | | 2 = 2+ |
| | | 3 = 3+ |
| | | NA = NA |
| | | . = Missing |

# 12.3 Identification of Patient's central pathology result

The classification of each result from IEO will be done before identifying which sample should be used for the central result.

# 12.3.1 Considerations

For the RoW patients the CRF data will be available for each accession number comprising;

Accession number, date sample taken, and time point either archival or surgical (see Blood/Tumour Samples (Screening)).

For the US patients CRF data is only available for archival samples and not necessarily all archival samples. The time point archival or surgical sample was taken will be available from IEO for the US patients as this is sent directly from NRG to IEO.

# 12.3.2 Identifying the central pathology result

This flow will be followed to programmatically identify the result to be used in the central pathology analysis.

# 1 Only one central time point result for an individual patient in the IEO data

- 1.1 No duplicates accession numbers for that result *Use this accession number to identify the result by central testing*
- 1.2 Duplicate accession number for that result Follow point 2 above (section 1.1) to identify the result by central testing

# 2 More than one central time point result for an individual patient in the IEO data

#### 2.1 RoW

# 2.1.1 Site know what time point they were randomised under

2.1.1.1 No duplicate accession numbers for that time point

Use this accession number to identify the result by central testing

2.1.1.2 Duplicate accession number for that time point

Follow point 2 above (section 1.1) to identify the result by central testing

# 2.1.2 Site don't know what time point they were randomised under

*Identify the earliest sample collection date reported on the CRF* 

2.1.2.1 No duplicate accession numbers for that date

*Use this accession number to identify the result by central testing* 

2.1.2.2 That date has duplicate accession numbers

Follow point 2 above (section 1.1) to identify the result by central testing

#### 2.2 US

# 2.2.1 Site know what time point they were randomised under

2.2.1.1 No duplicate accession numbers for that time point

Use this accession number to identify the result by central testing

2.2.1.2 Duplicate accession number for that time point

Follow point 2 above (section 1.1) to identify the result by central testing

#### 2.2.2 Site don't know what time point they were randomised under

*Use the archival time point sample* 

2.2.2.1 No duplicate accession numbers for the sample from the archival time point *Use this accession number to identify the result by central testing* 

2.2.2.2 The sample from the archival time point has duplicate accession numbers

*Follow point 2 above (section 1.1) to identify the result by central testing*